## Clinical Development

## AMN107 (Nilotinib, Tasigna®)

Study Number: CAMN107AIC05 / NCT01743989

A prospective, randomized, open-label, two-arm Phase III study to evaluate treatment-free remission (TFR) rate in patients with Philadelphia chromosome-positive CML after two different durations of consolidation treatment with nilotinib 300 mg BID

## **RAP Module 3- Detailed Statistical Methodology**

| Authors: | statistician |
|------------------|-------------------------------|
| Reviewers: | , Novartis study statistician |
| Document type: | RAP Addendum |
| Document status: | Final |
| Release date: | 16 Mar2021 |
| Number of pages: | 49 |

Property of Novartis


May not be used, divulged, published or otherwise disclosed without the consent of Novartis

Document History – Changes compared to previous version of RAP module 3.

| Version | Date | Changes |
|---|---|---|
| 1.0 | 13-Jan-2020 | Initial draft |
| 1.1 | 05-Mar 2020 | Draft v 1.1, Added analysis |
| 1.2 | 30-Mar-2020 | Format Changes |
| 1.3 | 06-Apr-2020 | Adding LSC sub-study abstract analysis |
| 1.4 | 01-July-2020 | Updating according to DR1 comments |
| 1.5 | 28-Sep-2020 | Adding LSC FAS definition |
| 1.6 | 06-Oct-2020 | Adding SSMC extra analysis |
| Pre- Final | 07-Oct-2020 | Finalize document |
| Final | 09-Oct-2020 | Minor cosmetics update and final version for CSR |
| Addendum | 04-Jan-2021 | Sensitivity analysis, excluding SDV (not done) involved visits KM analysis of PFS and TFS based on eCRF captured variable 'Progression to AP/BC' |
| Addendum<br>V1.1 | 29-Jan-2021 | Section 4.8, excluding Safety output Sensitivity analysis outputs not affected by the SDV record exclusion of specific visits, since they are based on Start and Stop dates independently of standard study visits: Duration of exposure, relative dose intensity, dose reduction/interruption of study drug treatment, Concomitant medication, AEs, TEAES, CVEs and Medical History. |
| Final | 16-03-2021 | Final version |

## **Table of contents**

| 1 Statistical methods planned in the protocol | | | | |
|---|---|---|---|---|
| 2 | Statis | tical and a | analytical plans | 8 |
| | 2.1 | Overvie | ew of study design | 8 |
| | 2.2 | Study ol | bjectives | 10 |
| | 2.3 | General | strategies of data presentation | 12 |
| | 2.4 | | nent windows, baseline and post-baseline definitions, missing da | |
| | | 2.4.1 | Time-windows | 12 |
| | | 2.4.2 | Assessment windows | 15 |
| | | 2.4.3 | Baseline and post-baseline definitions | 16 |
| | | 2.4.4 | Last contact date | 18 |
| | | 2.4.5 | Cut-off date | 18 |
| | | 2.4.6 | End of Study (EoS) visit | 18 |
| | 2.5 | Missing | data handling | |
| | 2.6 | Analysis | s proportions | 19 |
| | | 2.6.1 | Analysis of Molecular response proportions | 19 |
| | | 2.6.2 | Analysis of time-to-event endpoints | |
| | | 2.6.3 | Adjustment for covariates | |
| | 2.7 | Other de | efinitions | |
| | | 2.7.1 | Treatment periods and treatment emergent periods | 20 |
| | | 2.7.2 | TFR phase and emergent adverse events | |
| | | 2.7.3 | Cardiovascular risk factors | |
| | | 2.7.4 | Study medication | 22 |
| | | 2.7.5 | Duration of exposure | |
| | | 2.7.6 | Relative dose intensity | 23 |
| | | 2.7.7 | Molecular responses | 24 |
| | | 2.7.8 | Progression-free survival | 24 |
| | | 2.7.9 | Treatment-free survival | |
| | | 2.7.10 | Overall survival | 25 |
| | | 2.7.11 | LSC detected cases | 25 |
| 3 | Subje | ects and tre | eatments | 28 |
| | 3.1 | | on of analysis sets | |
| | 3.2 | | disposition and characteristics at screening | |
| | | 3.2.1 | Patient disposition | |
| | | 3 2 2 | Screen Failures | 31 |

| | | 3.2.3 | Study discontinuation | 31 |
|---|---|---|---|---|
| | | 3.2.4 | Demographics and baseline characteristics variables | 32 |
| | | 3.2.5 | Disease history | 34 |
| | | 3.2.6 | Medical history/current medical condition | 34 |
| | | 3.2.7 | Cardiovascular risk factors | 34 |
| | 3.3 | Prior ar | nd concomitant medications/non-drug therapies | 36 |
| | | 3.3.1 | Description of CV risk factors based on medical history, laboratory parameters and vital signs at baseline | |
| | 3.4 | Study n | nedication | |
| | | 3.4.1 | Duration of exposure | 38 |
| | | 3.4.2 | Relative dose intensity | 38 |
| | | 3.4.3 | Dose reduction and interruption | 38 |
| | | 3.4.4 | Dosage administration record | 38 |
| | 3.5 | Protoco | ol deviations | 38 |
| 4 | Effica | acy evalu | ation | 38 |
| | 4.1 | = | ılar response | |
| | 4.2 | Subgro | up definition | 39 |
| | | BCR-A | BL (IS) ratio at baseline | 39 |
| | | BCR-A | .BL (IS) ratio at Month 3 | 39 |
| | | Molecu | alar response up to Month 3 (suggested by SSMC members) | 39 |
| | | Halving | g time of BCR-ABL (IS) ratio | 40 |
| | | Time si | ince initial diagnosis of CML | 40 |
| | | Sokal r | isk group | 40 |
| | 4.3 | Kinetic | s of BCR-ABL(IS) transcript levels | 41 |
| | 4.4 | Progres | ssion free survival after entering the TFR phase | 41 |
| | 4.5 | Treatm | ent free survival after entering the TFR phase | 41 |
| | 4.6 | Overall | survival after Randomization | 41 |
| | 4.7 | Other e | fficacy assessments | 42 |
| | 4.8 | SDV se | ensitivity analysis | 42 |
| 5 | Pharr | nacokinet | tic evaluations | 43 |
| 6 | Safet | y evaluati | on | 43 |
| | 6.1 | Advers | e events | 43 |
| | 6.2 | Labora | tory abnormalities | 45 |
| | 6.3 | Vital si | gns | 46 |
| | 6.4 | Electro | cardiograms (ECGs) | 47 |
| | 6.5 | Echoca | rdiography (cardiac imaging) | 47 |

| | 6.6 | Survival Follow-up | 47 |
|---|-------|------------------------|----|
| | 6.7 | Safety Follow-up | 48 |
| | | LSC sub-study analysis | |
| 7 | Other | r topics | 49 |
| | | ole size calculation | |
| | | rences | |

#### List of abbreviations

ABL Abelson leukemia virus

AE Adverse Event

AESI Adverse Event of Special Interest

ALT Alanine aminotransferase/glutamic pyruvic transaminase/GPT

ANC Absolute Neutrophil Count

AP Accelerated phase

AST Aspartate aminotransferase/glutamic oxaloacetic transaminase/GOT

BC Blast Crisis

BCR-ABL oncoprotein product of BCR-ABL fusion gene

BID bis in diem/twice a day

CCyR Complete cytogenetic response
CHR Complete hematological response

CML Chronic myeloid leukemia

CP Chronic phase

eCRF Case Report/Record Form; the term CRF can be applied to either EDC or Paper

CSR Clinical study report

CTCAE NCI Common Terminology Criteria for Adverse Events

CV Cardiovascular

CVEs Cardiovascular events

DI Dose Intensity

DMC Data Monitoring Committee

ECG Electrocardiogram

ECOG Eastern Cooperative Oncology Group

EDC Electronic Data Capture

EoS End of Study

EUTOS European Treatment Outcome Study

FAS Full Analysis Set

FDA Food and Drug Administration (USA)

GFR Glomerular Filtration Rate

ICE Ischemic cerebrovascular events

IHD Ischemic heart disease
IS International scale
LLN Lower limit of normal

LVEF Left ventricular ejection fraction

MedDRA Medical dictionary for regulatory activities

MMR Major molecular response

MR Molecular response

MR<sup>40</sup> 4.0 log reduction on international scale (IS) MR<sup>45</sup> 4.5 log reduction on international scale (IS)

## Novartis Confidential Page 7 RAP Module 3 16-Mar-2021 (9:09) CAMN107AIC05

NEU Neutrophils

PAOD Peripheral arterial occlusive disease

PD Protocol deviation
PDI Planned Dose Intensity
PCR Polymerase chain reaction
Ph Philadelphia chromosome

Ph+ CML Philadelphia chromosome positive chronic myeloid leukemia

PFS Progression Free Survival

PPS Per Protocol Set
PT Preferred Term

RDI Relative Dose Intensity
SAE Serious adverse event
SDV Source Data Verification
SOC System Organ Class

SMQ Standardized MedDRA Query

TEAE Treatment Emergent Adverse Event

TFR Treatment free remission
TFS Treatment free survival
TKI Tyrosine kinase inhibitor
ULN Upper limit of normal
VAP Validation and planning

WBC White blood cell

## 1 Statistical methods planned in the protocol

This document contains details of the statistical methods which will be applied for the CSR analysis for the CAMN107AIC05 clinical trial.

The Primary objective of the CSR is to assess the optimal duration of consolidation treatment with nilotinib 300 mg BID in order that patients remain in treatment-free remission (≥MR4.0) without molecular relapse 12 months after entering the TFR phase

## 2 Statistical and analytical plans

The data will be analyzed by according to the data analysis section 10 of the study protocol which is available in Appendix 16.1.1 of the CSR. Important information is given in the following sections and details are provided, as applicable, in Appendix 16.1.9 of the CSR.

Analyses will be conducted on all enrolled patients (Full Analysis Set, excluding patients without major protocol deviation) and all their data will be used for the analyses.

Primary Endpoint analysis will be performed for both FAS and PPS (FAS, excluding patients without major protocol deviation.

Data will be summarized with respect to demographic and baseline characteristics and safety observations and measurements. Assessment of molecular response will also be summarized.

## 2.1 Overview of study design

The CAMN107AIC05 study is a prospective, randomized, open label, multicenter, two arm Phase III study that includes a 12-month induction phase, followed by a 12 or 24 months consolidation phase (dependent on randomization), and a 36 or 24 month TFR phase respectively, adding to 5 year study duration for the individual patient.

This study aims to assess the optimal duration of nilotinib 300 mg twice daily (BID, bis in die) consolidation treatment, in order that patients remain in TFR ( $\geq$  molecular response [MR]<sup>4.0</sup>) 12 months after starting the TFR phase of the study. Patients with chronic myeloid leukemia in chronic phase (CP CML) who have received 24 months of first line imatinib treatment, and who have failed to achieve the molecular response threshold for treatment cessation ( $\geq$ MR<sup>4.0</sup>) have a 50% greater chance of achieving this level of molecular response by switching to nilotinib; however the optimal duration of consolidation treatment with nilotinib to ensure the highest rate of patients remaining in  $\geq$ MR<sup>4.0</sup> after suspending treatment is not yet known. This study therefore aims to assess the potential impact of two durations of consolidation treatment with nilotinib, i.e. 12 months versus 24 months, on molecular relapse rate in the first 12 months of the TFR phase. Eligible patients are adults with a confirmed diagnosis of chronic phase Ph+ and/or BCR ABL+ CML who have been treated with first line imatinib for 2 calendar years or more and are in complete cytogenetic response (CCyR). Patients must not have achieved  $\geq$ MR<sup>4.0</sup> at study entry, as assessed/confirmed by a local or a EUTOS laboratory.

620 patients have been enrolled into the study and were treated with nilotinib 300 mg BID for 24 months. Following the 24 months of treatment, patients in sustained molecular response for at least the last 12 months will be randomized on a 1:1 basis to either:

- Suspend nilotinib treatment immediately and enter the TFR phase (Arm 1; the nilotinib 24 months treatment arm); or
- Continue nilotinib treatment for a further 12 months then suspend treatment and enter the TFR phase (Arm 2; the nilotinib 36 months treatment arm).

Treatment-phases will be labelled, using as reference time point Randomization visit, as:

- "Induction/consolidation treatment phase", for both treatment arms from the date of Informed consent until Randomization visit.
- ➤ "Post-randomization treatment phase (ARM2)" for the 12-month additional treatment for treatment arm 2, from the date of Randomization visit+ 1 day.

Patients not achieving a sustained molecular response at 24 months (and subsequently at 36 months if previously randomized to the treatment arm with 1 year additional consolidation) will exit the study and will be treated at the discretion of the Investigator according to standard practice. Information on survival, stem cell transplantation, and on the status of the patient's disease (i.e. disease progression to AP (accelerated phase)/BP (blastic phase) according to protocol definition, tyrosine kinase inhibitor (TKI) treatment) will be collected until death, or until 5 years from study entry, whichever comes first.

Patients relapsing during the TFR phase will enter the nilotinib re-treatment phase of the study and will be re-treated with the same dose of nilotinib as they were on before the TFR phase (i.e. the re-treatment dose will be nilotinib 300 mg BID or a lower dose of nilotinib if this was reduced in the consolidation phase before entering the TFR phase). These patients will remain on study until the completion of the 5 years study period.

Details on the visit schedules and assessments are reported in Section 7 of the study protocol.

Optional Leukemic Stem Cells ENESTPath sub-study:

The Stem cells ENESTPath sub-study aims to add the determination of Ph+ stem cells in bone marrow in those patients consenting to participate in this sub-study, at the following time points:

- a) At the screening visit, before starting nilotinib treatment
- b) After 24 months of nilotinib treatment at Visit 8
- c) After 36 months of nilotinib treatment, only in patients with 12 months additional of consolidation treatment (Arm 2) at Visit 204
- d) If the patient relapses during the TFR phase, before re-starting the treatment with nilotinib.

A 10 mL bone marrow sample is collected at each time point and sent to

for immunophenotype analysis, FACS (fluorescence activated cell sorting) cell purification, in situ hybridization, and RT-PCR. Measurement and quantification will be performed by flow cytometry in a bone marrow purified population of stem cells in order to detect the presence of leukemic Ph+ cells or BCR-ABL transcript levels (evaluated by fluorescent in situ hybridization [FISH] or RT-PCR).

## 2.2 Study objectives

The primary objective of the study is to assess the optimal duration of consolidation treatment with nilotinib 300 mg BID in order that patients remain in treatment free remission (TFR) with a molecular response of 4.0 or higher ( $\geq$ MR<sup>4.0</sup>) without molecular relapse 12 months after entering the TFR phase.

The secondary objectives of the study are:

- To evaluate the proportion of patients who are eligible to suspend nilotinib therapy by achieving and maintaining sustained ≥MR<sup>4.0</sup> for at least 12 months during consolidation phase with 300 mg BID nilotinib;
- To assess the kinetics of molecular response of patients during induction/consolidation treatment with 300 mg BID nilotinib;
- To assess the kinetics of molecular response in patients during the TFR phase of the study in both treatment arms;
- To assess progression-free survival (PFS) rate after randomization in both treatment arms;
- To assess treatment-free survival (TFS) rate after randomization in both treatment arms:
- To estimate overall survival (OS) rate after randomization in both treatment arms;
- To assess the safety profile of nilotinib during the induction/consolidation phase, the TFR phase, and during the re-treatment phase.

For those patients consenting to participate in the optional Stem cells ENESTPath substudy included in Amendment 1, the following objectives will be also evaluated:

- To evaluate the presence and amount of leukemic stem cells (LSC) and their progenitors in the bone marrow of all patients participating in this substudy before and after completing induction and first year of consolidation phase (at Visit 8);
- To evaluate if prolonging treatment period of consolidation with nilotinib (patients in Arm 2 versus patients in Arm 1) causes a reduction in the percentage of patients presenting LSC and progenitor cells in bone marrow at the end of the second year of consolidation phase;
- To perform an exploratory analysis in order to evaluate if relapse in patients during the TFR phase in either arm correlates with the presence of LSC and progenitor cells in bone marrow at the end of the consolidation phase.
- To check the correlation of the response after switch from Imatinib to Nilotinib with the persistence of LSCs in the blood.

Additionally, for LSC-sub-study data the following objectives were set:

- To evaluate LSC detected cases, by Prior Imatinib exposure, Major Molecular Response Age and Sokal score for Randomized vs Not Randomized.
- To evaluate the presence and amount of leukemic stem cells (LSC) in Arm 1m Arm 2, Randomized, Not Randomized and Total group of LSC detected cases.

| Objective | Endpoint | Analysis |
|---|---|---|
| To evaluate the presence and number of LSC and their progenitors in the bone marrow of all patients participating in this substudy before and after completing induction and first year of consolidation phase (at Visit 8). | Proportion of patients with presence of Ph+ LSC in bone marrow (CD34+/CD38+ progenitor cells, CD34+/CD38- stem cells, and Immunophenotypically aberrant CD34+ stem cells [the last ones only if detectable]) at screening and at Visit 8, and Immunophenotypically aberrant CD34- stem cells. | The percentage of patients presenting Ph+ LSC in bone marrow will be calculated at each time point and will be presented by descriptive statistics. |
| To evaluate whether prolonging the treatment period of consolidation with nilotinib (patients in Arm 2 versus patients in Arm 1) induces a reduction in the percentage of patients presenting LSC and progenitor cells in bone marrow at the end of the second year of the consolidation phase (Visit 204 for Arm 2 versus Visit 8 for Arm 1); | Proportion of patients with presence of Ph+ LSC in bone marrow (CD34+/CD38+ progenitor cells, CD34+/CD38- stem cells, and Immunophenotypically aberrant CD34+stem cells [the last ones only if detectable]) at the end of consolidation arm (Visit 8 for Arm 1 and Visit 204 for Arm 2) and Immunophenotypically aberrant CD34- stem cells. | Descriptive statistics. |
| To perform an exploratory analysis in order to evaluate whether relapse in patients during the TFR phase in either arm correlates with the presence of LSC and progenitor cells in bone marrow at the end of the consolidation phase and at the time of relapse during TFR. | Proportion of patients with or without molecular relapse in the first year of TFR in either arm by presence of LSC in bone marrow (CD34+/CD38+ progenitor cells, CD34+/CD38- stem cells, and CD34+/CD56+ aberrant stem cells [the last ones only if detectable]) at Visit 8 and at the time of relapse during TFR. | Descriptive statistics |

## 2.3 General strategies of data presentation

All categorical data will be summarized by frequencies and percentages, with the denominator being the total number of patients included in the analysis population, or the number of patients with available data (as specified in RAP Module 7).

Continuous data will be summarized with either standard descriptive statistics (i.e. the number of non-missing data, arithmetic mean, standard deviation, median, 25<sup>th</sup> and 75<sup>th</sup> percentiles, minimum and maximum), or will be collapsed into categorical data and summarized as categorical data.

Pre-randomization data will be presented for Arm1, Arm2, Not Randomized and Total.

Shells of the tables, listings and figures are described in Module 7 of the RAP.

# 2.4 Assessment windows, baseline and post-baseline definitions, missing data handling

#### 2.4.1 Time-windows

For analysis purposes, time-windows will be defined. The time-windows are defined so that there are no gaps between the planned assessments, i.e. every assessment, including additional unscheduled assessments, would be assigned to one specific time-point. If there is more than one assessment within the time-window, the last available assessment in that time-window will be used. For all time-windows after baseline, only values after first dose of study drug will be used.

- Pre randomization induction/consolidation phase (Arm1, Arm2 and Not Randomized), time-windows are defined as starts at first day of study treatment and ends with randomization date. For Not-Randomized patients V400 (End of Induction /Consolidation visit) will be used.
- For post-randomization consolidation phase (Arm 2 only), time-windows are defined as starting at randomization date + 1 day and ending with the last day of study treatment (12 months after first randomization + 1 day).
- For TFR phase, time-windows are defined based on first day of TFR phase (i.e. last day of study drug intake from induction/consolidation phase for Arm1 or last day of study drug intake from post-randomization consolidation phase for Arm2, as described in section 2.8.4 + 1 day).
- For re-treatment phase, time-windows are defined based on first day of re-treatment (i.e. first day of study drug intake when patient re-starts study drug as described in section 2.8.4). The following table shows the time-windows for the analyses of molecular response based on the planned assessment schedule.

Time-windows presented in Table 1 below are calculated using the following formula:

- When assessments are planned every month: Day ([xx-0.5]\*30.4375 + 1) Day ([xx+0.5]\*30.4375) where xx is the month of the visit
- When assessments are planned every 2 months: Day ([xx-1]\*30.4375 + 1) Day ([xx+1]\*30.4375) where xx is the month of the visit
- When assessments are planned every 3 months: Day ([xx-1.5]\*30.4375 + 1) Day ([xx+1.5]\*30.4375) where xx is the month of the visit
- For Day 1 and Week 6 time-window of re-treatment phase, Week 6 starts at Day ([6-3]\*7+1) and ends where Month 3 starts. Day 1 time-window ends the day before Week 6 starts (day 21).

Depending on the study phase, time-windows are defined based on reference start dates defined in section 2.4.2  below.

Table 1 Definition of time-windows for molecular response

| | Planned<br>visit | Study Day | Time- | window | Comment |
|---|---|---|---|---|---|
| Induction/Consolidation | | | | | |
| phase | Month 3 | Day 91 | 2 - | 136 | |
| | Month 6 | Day 183 | 137 - | 228 | |
| | Month 9 | Day 274 | 229 - | 319 | |
| | Month 12 | Day 365 | 320 - | 410 | Pre-Randomization |
| | Month 15 | Day 457 | 411 - | 502 | |
| | Month 18 | Day 548 | 503 - | 593 | |
| | Month 21 | Day 639 | 594 - | 684 | |
| | Month 24 | Day 731 | 685 - | 776 ^ | |
| | Month 27 <sup>\$</sup> | Day 822 | 777 - | 867 | |
| | Month 30 <sup>\$</sup> | Day 913 | 868 - | 959 | Post- Randomization |
| | Month 33 <sup>\$</sup> | Day 1004 | 960 - | 1050 | |
| | Month 36 <sup>\$</sup> | Day 1096 | 1051 - | 1141 ^ | |
| TFR phase | Month 1 | Day 30** | 1 - | 46# | |
| | Month 2 | Day 61 | 47 - | 76# | |
| | Month 3 | Day 91 | 77 - | 107# | |
| | Month 4 | Day 122 | 108 - | 137# | |
| | Month 5 | Day 152 | 138 - | 167# | |
| | Month 6 | Day 183 | 168 - | 213# | |
| | Month 8 | Day 244 | 214 - | 274# | |
| | Month 10 | Day 304 | 275 - | 335# | |
| | Month 12 | Day 365 | 336 - | 411# | |
| | Month 15 | Day 457 | 412 - | 502# | |
| | Month 18 | Day 548 | 503 - | 594 <sup>#</sup> | |

| | Month 21 | Day 639 | 595 - | 685# |
|--------------|--------------------------|----------|--------|-------|
| | Month 24 | Day 731 | 686 - | 776# |
| | Month 27 <sup>\$\$</sup> | Day 822 | 777 - | 867# |
| | Month 30 <sup>\$\$</sup> | Day 913 | 868 - | 959# |
| | Month 33 <sup>\$\$</sup> | Day 1004 | 960 - | 1050# |
| | Month 36 <sup>\$\$</sup> | Day 1096 | 1051 - | 1141# |
| Re-treatment | Day 1 | Day 1*** | 1 - | 21 |
| phase | Week 6 | Day 42 | 22 - | 67 |
| | Month 3 | Day 91 | 68 - | 137 |
| | Month 6 | Day 183 | 138 - | 228 |
| | Month 9 | Day 274 | 229 - | 320 |
| | Month 12 | Day 365 | 321 - | 411 |
| | Month 15 | Day 457 | 412 - | 502 |
| | Month 18 | Day 548 | 503 - | 594 |
| | Month 21 | Day 639 | 595 - | 685 |
| | Month 24 | Day 731 | 686 - | 776 |
| | Month 27 <sup>\$\$</sup> | Day 822 | 777 - | 867 |
| | Month 30 <sup>\$\$</sup> | Day 913 | 868 - | 959 |
| | Month 33 <sup>\$\$</sup> | Day 1004 | 960 - | 1050 |
| | Month 36 <sup>\$\$</sup> | Day 1096 | 1051 - | 1141 |

<sup>\*</sup> Reference start day is the first date of study drug exposure.

The presence and number of LSC and their progenitors in the bone marrow will be summarized for all enrolled patients participating in this sub-study before and after completing induction and the first year of the consolidation phase (at Visit 8 - Month 24), at the end of the second year of the consolidation phase (at Visit 204 - Month 36 for Arm 2).

Table 2 Definition of time-windows for LSC assessments

| | Text used in TLF | Planned visit | Study Day | Time-<br>window |
|---|---|---|---|---|
| Screening (Re-screening) | Baseline | Day 0 | Day 0 | <=1 |
| 12 <sup>th</sup> month of consolidation phase | Month 24 | V8-Month 24 | Day 731 | 685 -776 ^ |
| 24 <sup>th</sup> month of consolidation phase Arm 2 | Month 36 | V202- Month 36\$ | Day 1096 | 1051 -1141 @ |

<sup>^</sup>Randomization date or V400 for Not Randomized patients

<sup>\*\*</sup> Reference start day is the first day of TFR phase

<sup>\*\*\*</sup> Reference start day is the first day of re-treatment phase (i.e.

<sup>+ 1</sup> day after study drug intake when patient re-starts study drug).

 $<sup>^{\</sup>text{@}}$  Last day of study treatment (12 months after randomization date +1 day).

<sup>\$</sup> for patients in Arm 2 only.

<sup>#</sup> or last day before study drug re-start

Time window will be used, considering no gap should be allowed compared to the planned visit. It will permit to exclude visits performed long after the planned visit date.

Time-windows presented in Table 3 below are calculated using the following formula:

Assessments are planned every 3 months: Day ([xx-1.5]\*30.4375 + 1) – Day ([xx+1.5]\*30.4375) where xx is the month of the visit

Table 3 Definition of time-windows for Survival follow-up

| | Planned<br>visit | Study Day | Time | -window |
|--------------------|------------------|-----------|--------|---------|
| Survival follow-up | Month 3 | Day 91 | 2 - | 136 |
| | Month 6 | Day 183 | 137 - | 228 |
| | Month 9 | Day 274 | 229 - | 319 |
| | Month 12 | Day 365 | 320 - | 410 |
| | Month 15 | Day 457 | 411 - | 502 |
| | Month 18 | Day 548 | 503 - | 593 |
| | Month 21 | Day 639 | 594 - | 684 |
| | Month 24 | Day 731 | 685 - | 776 |
| | Month 27 | Day 822 | 777 - | 867 |
| | Month 30 | Day 913 | 868 - | 959 |
| | Month 33 | Day 1004 | 960 - | 1050 |
| | Month 36 | Day 1096 | 1051 - | 1141 |
| | Month 39 | Day 1187 | 1142 - | 1233 |
| | Month 42 | Day 1278 | 1234 - | 1325 |
| | Month 45 | Day 1370 | 1326 - | 1415 |
| | Month 48 | Day 1461 | 1416 - | 1507 |
| | Month 51 | Day 1552 | 1508 - | 1598 |
| | Month 54 | Day 1644 | 1599 - | 1690 |
| | Month 57 | Day 1735 | 1691 - | 1781 |
| | Month 60 | Day 1826 | 1782 - | 1873 |

<sup>\*</sup> Reference start day is the first day of survival follow-up.

#### 2.4.2 Assessment windows

Safety assessments will be performed at the following time-points:

- Screening (D-28 to D0)
- Baseline (D1)
- Every 3 months during the induction/consolidation phase
- End of Phase (EOP) visit

At each of the visit times stated above, peripheral blood will be taken for BCR-ABL RQ-PCR assessment (performed in EUTOS standardized laboratory) and hematological assessments.

Details on safety and efficacy assessments are reported in section 7 of the protocol.

For analysis purposes time-windows will be defined for the RQ-PCR, bone marrow, FISH test and biological assessments over the induction/consolidation phase.

The time-windows are defined so that there are no gaps between the planned assessments, i.e. every assessment, including additional unscheduled assessments, would be assigned to one specific time-point. If there is more than one assessment within the time-window, the last available assessment in that time-window will be used. For all time-windows after baseline, only values after first dose of study drug will be used. Time-windows are defined based on first study drug intake date (study day 1).

The following table shows the time-windows for the analyses of molecular response based on the planned assessment schedule.

Table 2 Time-window for analyses of RQ-PCR, bone marrow, FISH test and biological assessments

| Planned Assessment | Time-window |
|-----------------------------|------------------------------|
| Baseline | see definition in 2.5.2 |
| Month 3 – Day 91 | Day 2 – Day 136 |
| Month 6 – Day 182 | Day 137 – Day 228 |
| Month 9 – Day 273 | Day 229 – Day 319 |
| Month xx - Day (xx*30.4375) | Day ([xx-1.5]*30.4375 + 1) – |
| | Day ([xx+1.5]*30.4375) |

xx = Every 3 months until 24 months for Arm 1 and until 36 months for Arm 2.

#### 2.4.3 Baseline and post-baseline definitions

For all safety and efficacy evaluations the last available assessment before or on the date of start of study treatment is taken as the "baseline" assessment. If patients have no value as defined below, the baseline result will be missing. The study baseline is the same baseline as defined for the induction/consolidation phase. Except if it is specified differently, the term baseline will always refer to study baseline. The first day of start of study treatment is taken as "Day 1".

#### **Pre randomization Induction/consolidation phase:**

The last available assessment before or on the first day of nilotinib intake during induction/consolidation phase will be defined as the "baseline" assessment of the induction/consolidation phase.

The first day of start of study treatment is taken as "Day 1".

For adverse event, the day 1 will be considered as part of the post-baseline in the induction/consolidation phase.

Induction/consolidation phase end date corresponds to the last study drug administration date occurring before randomization/eligibility visit, or on the maximum date between:

- Randomization visit (date of visit 9) for Arm 1, visit 205 for Arm 2, and the
- End of induction/consolidation date (i.e. V400-EOP-ind/con date) for Not Randomized.

Pre-randomization induction/consolidation phase (CONS1) will be used for summary of AE. It corresponds to the 24 months of induction/consolidation phase (i.e. up to randomization) for arm 1 and arm 2.

#### Post-randomization consolidation for arm 2 (CONS2):

The randomization date + 1 day will correspond to the day 1 of this Post randomization consolidation phase. This sub-phase ends as defined for the end of induction/consolidation phase for arm 2.

#### **Treatment-free remission phase:**

The last available assessment before the first day of TFR phase (i.e. last day of nilotinib intake + 1 day) will be defined as the "baseline" assessment of the TFR phase.

The end date of TFR phase corresponds to the day of the first administration of re-treatment phase, defined as first study drug administration occurring after or on the maximum date between the end of TFR phase and the 1<sup>st</sup> visit from re treatment visit 301-RT day 1 date.

Any assessment occurring between the end date of induction/consolidation phase + 1 day and the end date of TFR will be considered as part of post-baseline in TFR phase.

#### **Re-treatment phase:**

The last available assessment before or on the end date of TFR phase (i.e. 1<sup>st</sup> day of re-treatment planned at visit V401-EOP-TFR) will be defined as the "baseline" assessment of the retreatment phase.

Start date of re-treatment phase corresponds to the end date of TFR phase + 1 day.

For the purpose of biochemistry/hematology shift tables, a "baseline" assessment will be used as mentioned above. If patients have no value as defined above, the baseline assessments will be missing.

For adverse event, the Day -1 of re-treatment phase (i.e. Day 1 of restart of nilotinib) will be considered as part of the post-baseline re-treatment phase.

Four study days will respectively be defined based on the reference start dates mentioned below:

- 1. Start of study drug exposure
- 2. Randomization date
- 3. Start of TFR phase date
- 4. Start of re-treatment phase date

Study days will be calculated from the reference start dates as follows:

• If the date of the event is on or after the reference date then: Study Day = (date of event – reference date) + 1. • If the date of the event is prior to the reference date then: Study Day = (date of event – reference date).

Study days will be used to show start/stop day of assessments and events in each phase as applicable.

#### 2.4.4 Last contact date

The last contact date will be derived as the maximum date when the patient is known to be alive. All dates from the databases will be checked (e.g. actual date of visit, laboratory assessment, AE, date of discontinuation, etc.) to determine the last contact date.

#### 2.4.5 Cut-off date

Cut-off date will be Last Patient Last Visit (LPLV) is scheduled.

## 2.4.6 End of Study (EoS) visit

End of study (EoS) visit where safety assessments if any will be collected, is planned when 5-years of study is completed. In case patient discontinued the study, EoS visit should be done immediately. When patient will complete the five years of study EoS visit will be performed without any time window.

## 2.5 Missing data handling

Throughout the study reasonable attempts will be made to limit the amount of missing data. However missing data will not be imputed, unless imputation is needed to perform specific analyses (e.g., for a dose administration record (DAR) with missing end date or end date after the cut-off date, the cut-off last contact date needs to be imputed as an end date to allow for calculation of treatment exposure duration and dose intensity). If it is required to impute an end date, the imputed date will be displayed and flagged in the appropriate listing, if produced. Imputation rules for missing dates (if applied) will be defined in the RAP Module 8 before the soft database lock.

The default rule for missing date imputation is the following:

- Day missing will be replaced by 15;
- Day & month missing will be replaced by 1July;
- No imputation if day, month and year are missing.

Imputed dates will not be displayed in listings except when required.

In the situation where the event date is partial or missing, the date will appear partial or missing in the listings, and study day, and any corresponding durations will be presented based on the imputations specified in the following paragraphs of this section.

For the analysis of PFS, time-to-first specific AE, overall survival (OS) and any time-to-first event, patients not meeting the event will be censored at the first date occurring between:

- the last contact date;
- the end of the applicable phase (if the event is specific to one phase);

- the cut-off date;
- date of death;

In case of missing PCR assessment, molecular response criteria will be imputed as follows: if no value exists in a time-window then the missing value will be imputed as a response if a response is observed on the last non-missing previous assessment and on the first next non-missing assessment (e.g. at Month 4, if a response is observed at the last previous assessment (i.e. Month 3) and at the next assessment (Month 5) then a response will be assumed at Month 4). If assessments are missing on two consecutive time-points, no imputation will be performed.

For the time-to-first specific AE analysis, patients not meeting the endpoint (=first occurrence of CVE) will be censored at the first date occurring between the (last treatment date + 30 days), the cut-off date and the date of death.

## 2.6 Analysis proportions

## 2.6.1 Analysis of Molecular response proportions

The proportion of successful TFR at 12 months, molecular responses or any other proportions will be calculated as the number of patients meeting the considered criterion divided by the number of patients in the analysis population (analysis populations will be specified in each section of this document).

Simple rates will be calculated by time window looking at all event between the start day and the end day of each time window. The number of patients at risk at the start point of time window will be used as denominator to compute the percentage of event in each time window.

Raw cumulative rates will be presented for each of the following phase:

- <u>Post-randomization consolidation phase for arm 2</u> using 1<sup>st</sup> study drug exposure date as starting point and each post-randomization timepoint after as stopping point: Day 822 (month 27), Day 913 (month 30), Day 1004 (month 33), Day 1096 (month 36), checking these stopping timepoint occurred before the start of the TFR phase.
- TFR phase using the start of TFR phase date as starting point and timepoint defined after: Day 30 (1 month), etc... repeat at each-time point every month, Day 183(month 6), etc... repeat at each-time point every two months, Day 365 (month 12), etc... repeat at each-time point every three months up to 36 month (Day 1096) for Arm 1 or up to 24 months (Day 721) for Arm 2 checking these stopping timepoint occurred before the start of re-treatment phase.
- Re-treatment phase using the start of re-treatment phase date as starting point and each timepoint after as stopping point: Day 42 (6 weeks), Day 91 (3 months), etc... repeat at each-time point every three months up to 36 months (Day 1096) for Arm 1 or up to 24 months (Day 721) for Arm 2.

The denominator to compute the cumulative rate in each phase above will be the number of patients in FAS with non missing start date of the phase.

## 2.6.2 Analysis of time-to-event endpoints

Time-to-event endpoints will be expressed in months. They will be analyzed using Kaplan-Meier estimates (product-limit estimates) that will be presented by treatment arm, together with a summary of the number (%) of events and censored patients. The associated statistics of the time-to-event endpoint will include median, first and third quartiles, and the corresponding two-sided 95% confidence intervals. Reference time point will be the randomization date + 1 day, or the date of entering in TFR phase, or date of entering in re-treatment phase, depending on the endpoint of interest. Censoring rules are provided in section 2.5.

#### 2.6.3 Adjustment for covariates

No covariates are defined in the study protocol.

#### 2.7 Other definitions

### 2.7.1 Treatment periods and treatment emergent periods

Per study design, patients are treated during the induction/consolidation phase (up to 24 months or 36 months depending on the randomization arm) and may also be treated again during the re-treatment phase (up to 36 months).

On-treatment period is defined from the first nilotinib dose intake up to the last intake of the considered phase.

Consequently, two treatment periods will be defined depending on the phase of the study.

Regarding treatment emergent abnormality or treatment emergent adverse event analysis, the treatment emergent period will be defined depending on the phase of the study:

- The treatment emergent period during pre-randomization induction/consolidation phase (for Arms 1 and 2) is defined as any event occurring between the first study drug dose intake, and the minimum date between last study drug dose intake + 30 days and the randomization date.
- The treatment emergent period during post-randomization consolidation phase (for Arm 2) is defined as any event occurring between the randomization date + 1 day and the minimum date between last nilotinib dose intake + 30 days and the start of TFR phase date.
- The treatment emergent period during re-treatment phase is defined as any event occurring between the start date of re-treatment phase and the last study drug dose intake during the re-treatment phase + 30 days.

#### 2.7.2 TFR phase and emergent adverse events

The emergent period during TFR phase is defined as the time between last study drug intake from (induction/consolidation phase for treatment Arm 1 or last study drug intake from post-randomization consolidation phase for treatment Arm 2, as described in section 2.8.4) + 1 day and end of trial / start of re-treatment.

All adverse events occurring during the TFR phase will be presented similar to the AEs occurring during post-randomization consolidation phase (Arm 2) or re-treatment phase (both treatment Arms). Since AEs occurring during TFR phase (i.e. not during treatment), they cannot be considered as TEAEs.

For example, TKI withdrawal syndrome" (e.g. muscle pain) may occur for the first period after the treatment discontinuation (i.e. during TFR). Although this Adverse Event technically can be considered as "treatment emergent AE", officially it is not, because the drug is no longer taken, so it will be included as an AE of Special Interest during TFR phase.

#### 2.7.3 Cardiovascular risk factors

Patients will be classified into 4 categories of cardiovascular (CV) risk factors at baseline according to the SCORE chart as described below:

#### 1. Very high risk:

Patients with any of the following criteria:

- At least one documented CV event (CVE) in their medical history as defined with the SMQ (Standardized MedDRA Query) and Preferred Term (PT) based on the last version of MedDRA associated to the following group of CVEs: CVEs (Ischemic heart disease (IHD)), CVEs (Peripheral arterial occlusive disease (PAOD)), CVEs (Ischemic cerebrovascular events (ICE)) and others CVEs. These groups will be defined based on a Novartis project-related document, the "Compound Case Retrieval Strategy" stored in CREDI under path: "Cabinets / CREDI Projects / A / AMN107A / Integrated Medical Safety". The updated version of this document effective at the time of the analysis will be used.
- Diabetes mellitus (type 1 or 2) history, as defined by LLTs based on the last version of MedDRA with one or more of the following CV risk factors: smoking history (current or ex-smoker), obesity (BMI at baseline>30 kg/m²), hypertension (severe or not) or dyslipidemia history (familial or not) as defined by PTs based on the last version of MedDRA, micro-albuminuria at baseline (20-200 mg/l)
- Severe chronic kidney disease, defined as a Glomerular Filtration Rate (GFR) <30 ml/min/1.73m<sup>2</sup> at baseline. GFR is measured by Cockcroft-Gault Creatinine Clearance rate as defined below:

```
GFR = [(140\text{-age})*weight (kg)*0.85 (for women)] / [Cr (umol/l)*0.814]
```

- A calculated HeartScore >=10% at baseline as defined by the European Guidelines on cardiovascular disease prevention in clinical practice (version 2012) and based on age, gender, smoking status, systolic blood pressure, total cholesterol and country.

#### 2. High risk:

Patients who did not meet any of the "Very high risk" criteria, and with any of the following criteria:

- Medical history of familial dyslipidemia or severe hypertension as defined by PTs based on the last version of MedDRA

- Diabetes mellitus (type 1 or 2) history as defined by LLTs, with no CV risk factor: non-smoker, BMI at baseline <=30 kg/m², no history of hypertension, no history of dyslipidemia, no micro-albuminuria (for diabetes mellitus patients with a missing BMI, missing smoker status or missing micro-albuminuria, the "Very high risk" category will be assumed)</li>
- Moderate chronic kidney disease defined as GFR>=30 ml/min/1.73m² and <=59 ml/min/1.73m²)</li>
- A calculated HeartScore >=5% and <10%

#### 3. Moderate risk:

Patients who did not meet any of the "Very high risk" or "High risk" criteria, and with a calculated HeartScore >=1% and <5%.

#### 4. Low risk:

Patients who did not meet any of the "Very high risk", "High risk" or "Moderate risk" criteria, and with a calculated HeartScore <1%.

If the HeartScore cannot be computed due to missing smoking history, age at baseline, gender, country, systolic blood pressure at baseline or total cholesterol at baseline then the CV category will be missing, except if other non-missing data classify the patient in the "Very high risk" category (i.e. document CVE, diabetes mellitus history with CV risk factor, GFR<30 ml/min/1.73m<sup>2</sup>).

If the GFR cannot be computed due to missing age at baseline, weight at baseline or creatinine at baseline then the CV category will be missing, except if other non-missing data classify the patient in the "Very high risk" category (i.e. document CVE, diabetes mellitus history with CV risk factor, HeartScore>=10%).

#### 2.7.4 Study medication

The investigational study drug used during the course of this trial is Nilotinib 300mg BID and will be supplied by Novartis for the duration of the trial.

Dosages may be adjusted for a number of reasons, see the protocol for details.

The number of patients who have dose reductions or interruptions, the number of dose reductions or interruptions, as well as their reasons, will be summarized. This will be done for all reductions or interruptions together and then summarized separately for reductions and for interruptions

#### 2.7.5 Duration of exposure

The following algorithm will be used to calculate the duration of nilotinib exposure per study phase:

• Duration of exposure (months) = (date of last study drug administration – date of first study drug administration + 1) / 30.4375

The duration includes the periods of temporary interruption.

The first administration for the exposure in the induction/consolidation phase is the first study drug administration taken from Drug Administration Recorded page of the CRF where daily dose administrated is not null/missing.

The last date of exposure in the induction/consolidation phase is defined as date of last study drug administration occurring before or on the maximum between:

- the date of Randomization for Arm1 (date of visit 9), visit 205 for Arm2)

#### And

- the end of induction/consolidation date (i.e. V400-EOP-ind/con date), including subjects Not Randomized.

The first administration of re-treatment phase is defined as first study drug administration occurring after or on the maximum date between the end of TFR phase and the 1<sup>st</sup> visit from retreatment visit 301-RT day 1 date.

First study drug administration for Arm 2 post-randomization consolidation phase starts at randomization date and ends at the last study drug administration date occurring before or on the TFR phase eligibility (i.e. date of visit 205 where eligibility is yes)

These dates of nilotinib administration are taken from Drug Administration Recorded page of the CRF where daily dose administrated is not null/missing.

The last date of exposure in the re-treatment phase is the last nilotinib administration of the study taken from Drug Administration Recorded (DAR) page of the CRF where daily dose administrated is not null/missing.

Duration of exposure will be analyzed separately for Pre-randomization induction/consolidation period, post-randomization consolidation period (ARM2) and re-treatment period.

### 2.7.6 Relative dose intensity

Relative dose intensity (RDI) is defined as follows: RDI = 100 \* DI (mg/day) / PDI (mg/day).

Planned dose intensity (PDI) is the assigned dose by unit of time planned to be given to patients as per protocol and is equal to 600 mg/day for nilotinib.

Dose intensity (DI) is defined as follows:

- DI (mg/day) = Cumulative dose (mg) / Duration of exposure (day).
- For patients who did not take any drug the DI is by definition equal to zero.

Cumulative dose is defined as the total dose taken by the patient during the study treatment exposure:

• Cumulative dose (mg) = sum of all rows on the dosage administration record of (actual dose \* (date of end of medication – date of start of medication + 1) (only '+1' if end date not the same as the start date of the next dose)).

Descriptive statistics of RDI as well as RDI by category will be presented. The categories of RDI presented will be 0 < 70%,  $\ge 70 < 90\%$ ,  $\ge 90 < 100\%$  and  $\ge 100\%$ .

The average daily dose will also be displayed, is defined as the DI: Cumulative dose (mg) / (date of end of medication – date of start of medication + 1) <math>(day).

Note that drug free days are included in the duration of exposure.

Listing for patients with dose administration records including start/stop dates, total dose and frequency, relative dose intensity and Discontinuation/Interruption along with the respective reason, will be presented.

#### 2.7.7 Molecular responses

- Molecular response 4.5 (MR<sup>4.5</sup>), defined as either detectable disease ≤0.0032% BCR to ABL(IS) ratio or undetectable disease in cDNA with ≥32,000 ABL transcripts. In case of undetectable disease, samples with a total of <32,000 ABL transcripts should be considered as not evaluable for MR<sup>4.5</sup>. Not evaluable samples will be classified as non-responder.
- Molecular response 4.0 (MR<sup>4.0</sup>), defined as either detectable disease ≤ 0.01% BCR to ABL(IS) ratio or undetectable disease in cDNA with ≥10,000 ABL transcripts. In case of undetectable disease, samples with a total of <10,000 ABL transcripts should be considered as not evaluable for MR<sup>4.0</sup>. Not evaluable samples will be classified as non-responder.
- Major molecular response (MMR), defined as a ≥ 3.0 log reduction in BCR-ABL transcripts compared to the standardized baseline or ≤ 0.1% BCR-ABL according to the international scale as measured by RQ-PCR.
- Relapse during TFR phase

As per protocol, relapse is defined as the loss of MMR, or the confirmed loss of MR4.0 (defined by three consecutive tests less than MR4.0 assessed at three consecutive visits according to the visit schedule of the TFR phase). If during the three consecutive tests, one of the tests shows loss of MMR, this patient will be declared as relapsing and will start the nilotinib re-treatment phase immediately even if the definition of confirmed loss of MR4.0 is not yet fulfilled. Molecular responses at specific time-windows will be used to define relapse, i.e. the last assessment of each time-window will be taken into account (see section ). In case of missing data, imputation of PCR assessment will be used as described in section 2.5.

#### 2.7.8 Progression-free survival

As per protocol, the progression of disease is defined as follows:

- Progression to accelerated phase (AP):
  - ≥ 15% blasts in peripheral blood or bone marrow aspirate, but <30% blasts in both peripheral blood and bone marrow aspirate
  - $\geq$  30% blasts plus promyelocytes in peripheral blood or bone marrow aspirate
  - $\geq$  20% basophils in peripheral blood
  - Thrombocytopenia ( $<100 \times 10^9/L$ ) that is unrelated to therapy

- Progression to blast crisis (BC):
  - $\geq$  30% blasts in peripheral blood or bone marrow aspirate
  - Appearance of extramedullary involvement other than hepato and/or splenomegaly proven by biopsy (i.e. chloroma)

For the purpose of analysis, failure of progression-free survival (PFS) will be defined as the earliest occurrence of progression to AP/BC (eCRF captured variable), or death for any cause after entering the TFR phase. The date of progression will be defined using the earliest assessment date among all criteria. In case of missing assessment date, the End of TFR phase visit date will be used.

If progression to AP/BC (eCRF captured variable) is not observed for the patient, patient will be censored as described in section 2.6.

#### 2.7.9 Treatment-free survival

According to the protocol for the purpose of the analysis, failure of treatment free survival (TFS), will be defined as the earliest occurrence of progression to AP/BC ((eCRF captured variable)), or loss of MMR, or confirmed loss of MR4.0, or re-start of nilotinib treatment for any reason, or death for any cause after entering the TFR phase. The date of failure will be defined using the earliest assessment date among all criteria. In case of missing assessment date, the End of TFR phase visit date will be used.

If failure of TFS is not observed for the patient, patient will be censored as described in section 2.6.

#### 2.7.10 Overall survival

As stated in the Protocol, one of the objectives of the CSR analysis is Overall survival, defined as the time from randomization to the time of death due to any cause after the date of Randomization. For randomized patients not known to have died on or before the cut-off date, survival time will be censored, at the date of last contact.

#### 2.7.11 LSC detected cases

LSC detected cases defined for Baseline, as the latest available valid evaluation between Screening and Re-screening), derived as follows:

- "LSC detected" when Ph+ for HIS, or PCR, or both regarding: CD34/38 +, or CD34/CD38 -, or Immunophenotypically aberrant CD34+ cells, or Immunophenotypically aberrant CD34 negative cells.
- "LSC not detected" in all other cases excluding missing and not evaluable observations. In general:
  - If any of the 8 evaluations is Positive then LSC detected: Yes
  - If there is NO Positive evaluation and at least one evaluation is Negative then LSC detected: **No**

If ALL 8 evaluations are Missing or Not Evaluable then **EXCLUDE**.

## Table 4 Table Example of LSC detection categories based on HIS and PCR results:

| | | <i>PH</i> + <i>i</i> | by HIS | | PH+ by PCR | | | | <u>LSC</u><br>detected |
|---|---|---|---|---|---|---|---|---|---|
| Subject | CD34+/<br>CD38+ | CD34+/<br>CD38- | Immuno-<br>phenotypical<br>ly aberrant<br>CD34+ cells | Immuno-<br>phenotypical<br>ly aberrant<br>CD34- cells | CD34+/<br>CD38+ | CD34+/<br>CD38- | Immuno-<br>phenotypical<br>ly aberrant<br>CD34+ cells | Immuno-<br>phenotypical<br>ly aberrant<br>CD34- cells | |
| 1 | Positive | Positive | Not<br>Evaluable | Not<br>Evaluable | Positive | Positive | Negative | Negative | Yes |
| 2 | Positive | Positive | Missing | Negative | Positive | Negative | Missing | Negative | Yes |
| 3 | Negative | Positive | Negative | Missing | Negative | Negative | Not<br>Evaluable | Missing | Yes |
| 4 | Negative | Negative | Negative | Missing | Positive | Missing | Negative | Not<br>Evaluable | Yes |
| 5 | Positive | Negative | Negative | Negative | Negative | Not<br>Evaluable | Missing | Negative | Yes |
| 6 | Negative | Negative | Positive | Negative | Negative | Negative | Not<br>Evaluable | Positive | Yes |
| 7 | Negative | Negative | Negative | Negative | Negative | Negative | Positive | Negative | Yes |
| 8 | Negative | Negative | Negative | Missing | Negative | Negative | Negative | Not<br>Evaluable | No |
| 9 | Negative | Negative | Negative | Missing | Missing | Negative | Missing | Negative | No |
| 10 | Negative | Negative | Negative | Negative | Missing | Not<br>Evaluable | Negative | Missing | No |
| 11 | Missing | Missing | Not<br>Evaluable | Missing | Missing | Missing | Missing | Missing | Excluded |
| 12 | Not<br>Evaluable | Not<br>Evaluable | Missing | Not<br>Evaluable | Not<br>Evaluable | Not<br>Evaluable | Not<br>Evaluable | Not<br>Evaluable | Excluded |

## 3 Subjects and treatments

### 3.1 Definition of analysis sets

**Enrolled population**: All enrolled subjects.

**Randomized Set:** All randomized patients. This analysis set will only be used for major protocol deviation listing and overall survival after randomization.

#### **Full Analysis Set**

The Full Analysis Set (FAS) will include all enrolled subjects, excluding patients with PD severity codes (0, 8).

**Safety population (SAF)**: The safety population consists of all subjects in the FAS who receive at least one dose of study medication, excluding patients with PD severity code 5. This set will be named "all treated patients" for the purpose of efficacy and safety analysis

**Survival Follow-up**: All enrolled subjects who were followed for progression and/or survival after premature withdrawal from any phase.

**Per-Protocol Set (PPS)**: The PPS consists of a subset of the patients in the FAS who are compliant with requirements of the clinical study protocol. Compliant with requirements of the clinical study protocol includes patients without major PD with severity code 1.

LSC sub-study Full Analysis Set (LSC FAS): The LSC FAS consists of a subset of the patients in the FAS who are also part of PPS and SAF, i.e. excluding patients with PD severity codes (0, 1, 5, 8).

Protocol deviations (PD), will be specified prior to database lock.

Criteria defining PD and their corresponding severity codes are provided in the Module 3 of the Validation and planning document (VAP version 8).

Major protocol deviations defined for CSR are described as below:

**Table 3 Protocol Deviations** 

| Analysis Set | Severity<br>Code | PD severity codes leading to exclusion from analysis set |
|---|---|---|
| FAS, PPS | 0 | Exclude from all efficacy analysis |
| SAF | 5 | Exclude from all safety analysis |
| FAS, SAF,<br>PPS | 8 | Exclude from all analysis |
| PPS | 1 | Exclude from Per-Protocol analysis |

For CSR analysis, all subjects from FAS will be included in the analyses. The primary analysis will be repeated on the PPS.

### 3.2 Patient disposition and characteristics at screening

#### 3.2.1 Patient disposition

The number of patients treated in induction/consolidation phase will be summarized as applicable during the study progress, as well as the number of patients who discontinued the induction/consolidation phase, along with the primary reason for discontinuation.

The summary of patients' disposition will be presented overall and also by year-phase combination: Induction-Consolidation 1st year, Induction-Consolidation 2nd year (prerandomization consolidation) and 3rd year of treatment (post-randomization consolidation) for ARM 2 patients only.

Number of patients not randomized, along with the respective reason, based on Molecular response criteria will be summarized. Considering that the standard criterion was defined as having 4 out of 5 quarterly assessments of ≥MR4.0 by a (EUTOS) standardized laboratory over the last 12 months AND the last assessment before randomization is at least MR4.0, the following categories for Not Randomized patients will be presented:

- o Patient with last assessment < MR4.0
- o Patient with <4 times, out of 5 MR4.0
  - Patient with 0 out of 5 times MR4.0
  - Patient with 1 out of 5 times MR4.0
  - Patient with 2 out of 5 times MR4.0
  - Patient with 3 out of 5 times MR4.0
- o Patient with 4 out of 5 times MR4.0 but last assessment < MR4.0
- o Patient with <4 times, out of 5 MR4.0 and last assessment MR4.0
- Other reason not related to Molecular response, including: AE, ICF withdrew, PD, lost to follow up, death, etc.

The following information will also be reported:

Number (percentage) of patients who are:

- Randomized
- Arm 1 Nilotinib 24-month treatment / Arm 2 Nilotinib 36-month treatment
  - o Patients completed the consolidation phase
  - o Patients discontinued before TFR phase
  - o Patients entered in the TFR phase
  - Patients who completed the TFR phase \*
  - o Patients in the TFR phase with 6 months (i.e. 213 days) without relapse
  - o Patients in the TFR phase with 12 months (i.e. 411 days) without relapse
    - entering in survival follow-up period
    - completing the survival follow-up and the 5 years study period
    - completing the survival follow-up before the 5 years study period

- discontinued from the study without survival follow-up
- o Patients discontinued TFR phase without entering re-treatment phase
  - entering in survival follow-up period
  - completing the survival follow-up and the 5 years study period
  - completing the survival follow-up before the 5 years study period
  - discontinued from the study without survival follow-up
- o Patients entered in the re-treatment phase
- Patients discontinued the re-treatment phase
  - entering in survival follow-up period
  - completing the survival follow-up and the 5 years study period
  - completing the survival follow-up before the 5 years study period
  - discontinued from the study without survival follow-up
- o Patients who completed the re-treatment

The duration of study will be described as: (date of last contact – date of informed consent + 1)/30.4375.

Percentages will be computed per arm over the number of patients randomized, over the patients entered in TFR phase, over the patient discontinued TFR, over the patient entered in retreatment phase or over the patient discontinued the re-treatment phase as mentioned in the TLF shells.

• Number of patients with no major deviation from protocol, due to which patients are excluded from safety or efficacy analysis (for analysis using Per Protocol Set).

Note that for Arm 1 TFR phase can be up to 36 months and re-treatment phase can be up 36 months, while for Arm 2 TFR phase can be up to 24 months and re-treatment phase can be up 24 months.

The number of patients in TFR phase at each month before Month 6, at every 2 months from Month 6 until Month 12 and every 3 months after Month 12, will be summarized. The number of patients in re-treatment phase will also be summarized at Week 6, Month 3 and every 3 months after.

A listing of all patients will be provided including the date of enrolment, the date of first and last study medication, the date of last contact, did the subject completed the study, discontinued the study and reason for discontinuation.

A listing will include details on subjects' last known date of study medication intake and whether the patient is followed up for survival, stem cell transplantation and disease progression to AP/BP from study entry and death date if applicable.

<sup>\*</sup>Completion of TFR phase is 36 months for arm 1 and 24 months for arm 2.

In addition, for patients participating in the LSC sub-study the following information will also be reported:

- Number of enrolled patients in the LSC sub-study (signed ICF for LSC sub-study).
- Number of enrolled patients in the LSC sub-study who received at least one dose of nilotinib
- Number of randomized patients per center and per country Percentages will be computed over the number of patients enrolled in the in the LSC sub-study
- Number of randomized patients:
  - In Arm 1: Percentages will be computed over the number of patients randomized in Arm1, as mentioned in the TLF shells.
  - In Arm 2: Percentages will be computed over the number of patients randomized in Arm 2 as mentioned in the TLF shells. Number of patients with no major deviation from protocol, due to which patients are excluded from safety or efficacy analysis.

#### 3.2.2 **Screen Failures**

Patients not fulfilling inclusion/ exclusion criteria at Baseline (Latest visit between Screening and Re-Screening), a table presenting the Reason of Screen failure as specific text presenting Inclusion- Exclusion Criteria depending on Protocol version will be created.

A listing presenting all Screen Failures including number and specific text on Inclusion/ Exclusion Criteria along with the respective Protocol version number, will be created.

#### 3.2.3 Study discontinuation

The following information will be reported in the FAS per treatment arm and overall:

Number (percentage) of patients discontinued along with primary reason for discontinuation:

- At any time point after randomization
- Before entering TFR
- After entering the TFR phase
- After entering re-treatment phase

A listing of patients who discontinued will be provided per study phase (induction phase, prerandomization consolidation phase, post-randomization consolidation phase (arm 2), TFR phase and re-treatment phase), including the reason for discontinuation, the date of end of phase, the last known date the patient took the treatment, and whether the patient continues to be followed for survival.

A listing of patients relapsing during TFR phase, but not entered immediately or never entered re-treatment phase, will be provided.

Study discontinuation and Protocol Deviation Listings will be created.

### 3.2.4 Demographics and baseline characteristics variables

Demographics and baseline characteristics will be summarized using the FAS per treatment arm, per randomization status (Randomized vs Not Randomized) and overall:

- Age at baseline visit in years, both numeric and categorical ( $<65 \& \ge 65$ )
- Gender (male, female)
  - o If female, child bearing potential (able to bear children, premenarche, post menopausal, sterile of child bearing age)
- Race (Caucasian, Black, Asian, Native American, North African descent, unknown, other)
- Eastern Cooperative Oncology Group (ECOG) performance status (World Health Organization (WHO))
- BMI (kg/m²) both numeric and categorical (very severely underweight (less than 15.0), severely underweight ( $\geq$ 15.0 <16.0), underweight ( $\geq$ 16.0 <18.5), normal ( $\geq$ 18.5 <25.0), overweight ( $\geq$ 25.0 <30.0), obese class I ( $\geq$ 30.0 <35.0), obese class II ( $\geq$ 35.0 <40.0) and obese class III ( $\geq$ 40.0))
- Smoking history (no, yes, ex-smoker)
  - If ex-smoker: duration (months) since stopped smoking, calculated as (date of screening visit date stopped smoking + 1) / 30.4375. Imputation of missing or partial dates will be handled as described in section 2.5.
  - o If yes or ex-smoker, use of tobacco products in the past 1 month (cigarettes, cigars, tobacco, other)
- Family history: presence of family diabetes, hypertension, dyslipidemia, cardiac events, cerebrovascular events and peripheral arterial disease.

Comparison between Randomized and No Randomized group will be done for Demographics and baseline characteristics, History of prior Imatinib therapy, Cardiovascular risk factors,

using: Pearson's Chi-square test p-value, or Fisher's exact test in case we have one or more frequencies in the cross-tabulation MR<sup>4.0</sup> Yes/No\*Randomized/Not Randomized, less than 5 for categorical variables, to check correlation between MR<sup>4.0</sup> and Randomization group.

For numeric variables, Independent t-test for mean (using "Equal" variances or "Unequal" variances depending on Variance test result) and Median test for median will be used to test for differences between Randomized and Not Randomized group.

- Listings will also be provided to display demographic data, as well as family history (from eCRF page).

## \*\*Sample pseudo SAS code for Pearson's and Fisher's Chi-square test for Categorical cross-tabulations\*

## \*Pearson chi-square test; ods trace on/listing; ods output ChiSq=pchisq; proc freq data=DATA; tables VAR\*trtg/chisq; run; ods trace off;

\*Keep prob where Statistic="Chi-Square";

#### \*Fisher's exact test;

ods trace on/listing; ods output FishersExact=fishert; proc freq data=DATA; tables VAR\*trtg/fisher; run; ods trace off;

\*Keep nValue1 where Name1="XP2 FISH";

### \*2 Independent samples t-test;

ods trace on/listing; ods output TTests=ttest; Equality=eqv;proc ttest data=data; class trtg; var age; run; ods trace off;

 $In\ probf >= 0.05\ in\ EQV\ dataset\ then\ in\ the\ ttest\ keep\ probt\ for\ Variances='Equal';$   $In\ probf\ < 0.05\ in\ EQV\ dataset\ then\ in\ the\ ttest\ keep\ probt\ for\ Variances='Unequal';$ 

#### \*Median test;

ods trace on/listing; ods output MedianTest=medt; proc nparlway data= data; class trtg; var var; run; ods trace off;

\*nValue1 where Name1='P2 MED';

### 3.2.5 Disease history

Disease History will be described in the FAS per treatment arm and overall as follows:

- Time since initial diagnosis (months) calculated as (date of the screening visit date of initial diagnosis) / 30.4375. Imputation of missing or partial dates will be handled as described in section 2.6.
- Peripheral blood blasts % at diagnosis
- PB eosinophils % at diagnosis
- PB basophils % at diagnosis
- Platelets at diagnosis (10<sup>9</sup>L)
- Spleen size at diagnosis (cm)
- Extramedullary involvement other than hepato and/or splenomegaly (yes, no)
- Sokal score at diagnosis, both continuous and categorical (low risk (<0.8), intermediate risk ( $\ge 0.8 \le 1.2$ ) and high risk (>1.2))
- Euro (Hasford) score at diagnosis, both continuous and categorical (low risk (≤780), intermediate risk (>780-≤ 1480) and high risk (>1480))
- EUTOS score at diagnosis, both continuous and categorical (high risk (>87) and low risk (≤87))
- Previous progression to AP/BP (yes, no)
- Attempt to stop treatment with Imatinib (yes, no)
- Molecular response at screening (BCR-ABL<sup>IS</sup> > 1%, BCR-ABL<sup>IS</sup> > 0.1  $\leq$  1%, > 1%, BCR ABL<sup>IS</sup> > 0.01  $\leq$  0.1%, BCR-ABL<sup>IS</sup>  $\leq$  0.01%, Undetectable BCR-ABL)

A listing will also be provided to display disease history.

### 3.2.6 Medical history/current medical condition

Medical history/current medical condition will be summarized in the FAS per treatment arm and overall by MedDRA System Organ Class (SOC) and Preferred Term (PT). A patient will be counted only once within a given SOC and within a given PT, even if he had several records.

A listing will also be provided, including MedDRA SOC and PT, verbatim, date of diagnosis/surgery, and whether the condition is still ongoing.

#### 3.2.7 Cardiovascular risk factors

Cardiovascular risk factors will be described with the following categories: very high risk, high risk, moderate risk and low risk, per treatment arm and overall.

Also, based on their medical history, the number and percentage of patients showing the following CV risk factors will be described:

- CVEs (IHD: Ischemic heart disease)

- CVEs (PAOD: Peripheral arterial occlusive disease),
- CVEs (ICE: Ischemic cerebrovascular events)
- CVEs (Others)
- Hypercholesterolemia
- Hypertension
- Diabetes
- At least one CV medical history

In addition, the number and percentage of patients meeting the following criteria based on laboratory parameters and vital signs at baseline will be described:

- Fasting glucose at baseline:
  - 5.6 6.9 mmol/L
  - >6.9 mmol/L
- Total cholesterol at baseline (> 5.2 mmol/L)
- LDL cholesterol at baseline (> 3.3 mmol/L)
- HDL cholesterol at baseline (< 1.3 mmol/L)
- Triglycerides at baseline (> 1.7 mmol/L)
- At least one risk factor between high total cholesterol, high LDL, low HDL, and high triglycerides
- Blood pressure at baseline (systolic blood pressure > 140mmHg or diastolic blood pressure > 90 mmHg) by treatment Arm and treatment phase:
  - ➤ Arm1
    - TFR
    - Re-treatment phase
  - ➤ Arm2
    - Post-randomization consolidation phase
    - TFR
    - Re-treatment phase

Listing will be provided to display CV risk factors with medical history, laboratory parameters and vital signs at baseline.

## 3.3 Prior and concomitant medications/non-drug therapies

Prior medications are defined as medications which started and stopped before the date of first nilotinib intake. Medications ongoing at the date of first nilotinib intake, as well as medications started after the date of first nilotinib intake, are defined as concomitant medications. In addition, concomitant medications will be classified by study phase (induction/consolidation, TFR, retreatment phases) depending on whether their start dates is before or after the reference start dates defined in section 2.5.

- Prior medication: start date of medication before the date of first nilotinib intake.
- Concomitant medication during induction/consolidation phase: start date of concomitant medication equal or after the date of first nilotinib intake, and before the first day of TFR phase.
- Concomitant medication during TFR phase: start date of concomitant medication equal or after the first day of TFR phase and before the end date of TFR phase.
- Concomitant medication during re-treatment phase: start date of concomitant medication equal or after the end date of TFR phase (first day of nilotinib administration in re-treatment phase).

In order to define prior/concomitant medications, missing or partial start and stop dates will be imputed as described in section 2.5.

A focus will be given on prior Imatinib, with the history of prior exposure summarized by both summary statistics and categorical frequencies (< 2 years,  $\geq$  2 years - < 5 years,  $\geq$  5 years). Duration of prior Imatinib exposure (months) will be calculated as (end date of prior imatinib intake – start date of prior imatinib intake + 1) / 30.4375.

Concomitant medications will be described per treatment arm and overall by therapeutic class and PT during induction/consolidation and TFR phase, and during the re-treatment phase in the subset of patients entering the re-treatment phase.

Listings of prior and concomitant medications will be provided, including ATC level 2, PT, verbatim, indication, start and stop dates, dose, frequency and route of administration. A specific listing will be provided for prior antineoplastic therapies, also including the therapy type and reason for discontination of therapy.

Prohibited medication will be presented in Listings for Full Analysis Set patients, including all necessary basci information (Country/Center/ patient number, age/sec/race) and Preferred term, ATC level 2 code, Indication, Start/End dates, phase of administratin, route of administration along with Dose and Frequency.

# 3.3.1 Description of CV risk factors based on medical history, laboratory parameters and vital signs at baseline

Based on their medical history, the number and percentage of patients showing the following CV risk factors will be described per treatment arm and overall:

- CVEs (IHD: Ischemic heart disease)
- CVEs (PAOD: Peripheral arterial occlusive disease),
- CVEs (ICE: Ischemic cerebrovascular events)
- CVEs (Others)
- Hypercholesterolemia
- Hypertension
- Diabetes
- At least one CV medical history

In addition, the number and percentage of patients meeting the following criteria based on laboratory parameters and vital signs at baseline will be described:

- Fasting glucose at baseline:
  - 5.6 6.9 mmol/L
  - 6.9 mmol/L
- Total cholesterol at baseline (> 5.2 mmol/L)
- LDL cholesterol at baseline (> 3.3 mmol/L)
- HDL cholesterol at baseline (<1.3 mmol/L)
- Triglycerides at baseline (> 1.7 mmol/L)
- At least one risk factor between high total cholesterol, high LDL, low HDL, and high triglycerides
- Blood pressure at baseline (systolic blood pressure > 140mmHg or diastolic blood pressure >90 mmHg)

Listing will be provided to display CV risk factors with medical history, laboratory parameters and vital signs at baseline.

## 3.4 Study medication

During pre-randomization induction/consolidation phase, both treatment arm patients will receive nilotinib for 24 months.

After randomization, there are two phases of the study when patients will take nilotinib:

- During the consolidation phase for Arm 2 (12 additional months of treatment before entering TFR phase)
- During the re-treatment phase in case of relapse during TFR phase (up to 24 or 36 months of treatment depending on the randomization arm)

The exposure to study medication will be described separately for the 2 above phases by treatment arm.

#### 3.4.1 Duration of exposure

The duration of exposure in months, will be described as a continuous variable and per category (< 6, >=6 - <12, >=12 - <18, >=18 - <24, >=24 - <30, >=30 - <36, >=36), by treatment arm and phase of study: pre-randomization induction/consolidation phase, consolidation (for Arm 2) and re-treatment phase.

#### 3.4.2 Relative dose intensity

Descriptive statistics of RDI will be presented, as well as RDI categories: 0 < 70%,  $\ge 70 < 90\%$ ,  $\ge 90 < 100\%$  and  $\ge 100\%$ .

The average daily dose will also be displayed, and is defined as the DI:

DI = Cumulative dose (mg) / (date of end of medication – date of start of medication + 1) (day).

Drug free days will be included in the duration of exposure.

#### 3.4.3 Dose reduction and interruption

The number of dose reductions or interruptions per patient will be summarized using the following categories: 0, 1, 2-3, more than 3 reductions/interruptions.

The number of patients with at least one dose reduction/interruption will be summarized, as well as the reason for reduction/interruption.

#### 3.4.4 Dosage administration record

A listing of the dosage administration records in induction/consolidation phase and in retreatment phase will be provided, including the dose administered, frequency, start and stop dates, whether the dose was changed/interrupted/permanently discontinued and the reason.

#### 3.5 Protocol deviations

The number of patients with any protocol deviations due to which patients are excluded from safety or efficacy analysis will be described in a frequency table based on the Enrolled patients. A listing describing the patients with any major protocol deviations due to which patients are excluded from safety or efficacy analysis will be provided.

# 4 Efficacy evaluation

All efficacy analyses will be performed on the set of Full Analysis Set, per treatment arm (including Not Randomized patients (as applicable) and Randomized as separate columns) and overall.

#### 4.1 Molecular response

Primary endpoint defined as MR<sup>4.0</sup> at 12 months of TFR, will be presented and compared for Arm1 vs Arm2, using Pearson's Chi-square test p-value, or Fisher's exact test in case we have one or more frequencies in the cross-tabulation MR<sup>4.0</sup> Yes/No\*Randomized/Not Randomized, less than 5 for subset of FAS entering the TFR phase, PPS, FAS and PPS.

The cumulative incidence of patients achieving MMR, MR<sup>4.0</sup> or MR<sup>4.5</sup> at selected time points of post-randomization (ARM2 patients) and re-treatment phase, as well as cumulative incidence of patients' loss of MMR, MR<sup>4.0</sup> or MR<sup>4.5</sup> during TFR phase as described in section 2.7.1 will be reported.

Note that for loss of MR4.5 population will be restricted to patients achieving MR4.5 as only MMR and MR4.0 are expected to be achieved for all patients eligible for TFR phase.

In addition, the proportions of MMR, MR<sup>4.0</sup> and MR<sup>4.5</sup> will be described based on time-windows described in section 2.4 (i.e. the last value of the time-window will be displayed).

The raw cumulative incidence of response will also be graphically displayed over time.

Listings presenting the BCR-ABL(IS) ratio, the total number of ABL copies, and the molecular response(s) for each phase will be provided.

#### 4.2 Subgroup definition

#### BCR-ABL (IS) ratio at baseline

The following subgroups will be defined based on the BCR-ABL (IS) levels at Baseline:

- BCR-ABL(IS) ratio >1%
- BCR-ABL(IS) ratio > 0.1%  $\le 1\%$
- BCR-ABL(IS) ratio > 0.01%  $\le 0.1\%$
- BCR-ABL(IS) ratio  $\leq 0.01\%$  (0% excluded)
- Undetectable BCR-ABL (when BCR-ABL(IS) ratio = 0 and the total number of ABL copies>10,000)

#### BCR-ABL (IS) ratio at Month 3

The following subgroups will be defined based on the BCR-ABL (IS) levels at Month 3 (i.e. last non missing assessment of the corresponding time-window):

- BCR-ABL (IS) ratio at Month  $3 \le 0.005\%$  (non missing value lower or equal to 0.005)
- BCR-ABL (IS) ratio at Month 3 > 0.005%

#### Molecular response up to Month 3 (suggested by SSMC members)

The following subgroups will be defined based on the derived molecular response up to

- Month 3:
  - Molecular response 4.0 up to Month 3
  - Molecular response 4.5 up to Month 3

#### Halving time of BCR-ABL (IS) ratio

The following subgroups will be defined based on the halving time, i.e. the time to reach a decrease in BCR-ABL (IS) ratio levels of at least 50% from baseline:

- Halving time <= 3 months (91 Days)
- Halving time > 3 months (91 Days)

The halving time will be computed as follows:

- Halving time = -d \* log(2)/[log(b)-log(a)]

#### where:

- a, is the Baseline BCR-ABL (IS) ratio value
- b, is the last Month 3 BCR-ABL (IS) ratio value
- d, is the actual treatment time in days over the two measurements

## Suboptimal response

Suboptimal response for patients who prematurely discontinued induction/consolidation phase using the following criteria:

- loss of CHR n (%)
- loss of CCyR n (%)
- loss of MMR n (%)
- no MMR up to Month 24 n (%)

Will be summarized in tables for Pre-randomization and Post-randomization (ARM2) phase.

## Time since initial diagnosis of CML

The following subgroups will be defined based on Time since initial diagnosis of CML:

- <2 years
- 2 to 4 years
- 4 to 6 years
- 6 to 8 years
- 8 to 10 years
- 10 to 12 years
- $\rightarrow$  = 12 years

#### Sokal risk group

The following subgroups will be defined based on Sokal risk category:

- Low risk (<0.8)
- Intermediate risk ( $\geq =0.8 \leq 1.2$ )
- High risk (>1.2)

## 4.3 Kinetics of BCR-ABL(IS) transcript levels

Descriptive statistics of BCR-ABL (IS) ratio will be provided at selected time points based on time-windows described in section **** (i.e. the last value of the time-window will be displayed):

- For Pre-randomization phase (Arm1, Arm2): Baseline (Month 0) and every 3 months until Month 24.
- For treatment phase (Arm 2): Month 24 (Randomization), and every 3 months until Month 36.
- For TFR phase: every month until Month 6, every 2 months until Month 12, and every 3 months until Month 24 or 36 depending on the randomization arm. This will be described per treatment arm and overall.
- For re-treatment phase: Day 1, Week 6, Month 3 and every 3 months until Month 36. This will be described in the subset of patients entering the re-treatment phase.

Listings presenting the BCR-ABL(IS) ratio, the total number of ABL copies, and the molecular response(s) will be provided for all patients at each phase.

#### 4.4 Progression free survival after entering the TFR phase

The evaluation of PFS after entering the TFR phase will be estimated in the two treatment arms of the FAS population sub-set entering the TFR phase, using Kaplan-Meier analysis. Summary statistics from the Kaplan-Meier distributions will be determined, as well as the proportions of patients remaining progression-free at 6, 12, 18, 24, 30 and 36 months after entered the TFR phase. The incidence of event will be graphically displayed.

A listing of the assessment of PFS will be provided.

#### 4.5 Treatment free survival after entering the TFR phase

The evaluation of TFS after entering the TFR phase will be estimated in the two treatment arms of the FAS population sub-set entering the TFR phase, using Kaplan-Meier analysis. Summary statistics from the Kaplan-Meier distributions will be determined, as well as the proportions of patients remaining treatment-free at 6, 12, 18, 24, 30 and 36 months after entered the TFR phase. The incidence of event will be graphically displayed.

A listing of the assessment of TFS will be provided.

#### 4.6 Overall survival after Randomization

The evaluation of OS after Randomization will be estimated in the two treatment arms of the FAS population sub-set Randomized, using Kaplan-Meier analysis. Summary statistics from the Kaplan-Meier distributions will be determined, as well as the proportions of patients survived at 6, 12, 18, 24, 30 and 36 months after entered the Randomization. The incidence of event will be graphically displayed.

A listing of the assessment of OS will be provided.

#### \*Sample pseudo SAS code for Kaplan Meier time to Event analysis;

#### \*Sample SAS code for Primary Efficacy;

Please check Pearson's and Fisher's exact test in section 3.2.4

## 4.7 Other efficacy assessments

Listings of bone marrow analysis, mutational analysis and extramedullary involvement will be provided for patients who underwent these assessments during the course of the study.

Listings presenting the Bone Marrow efficacy related data: Type of bone marrow sample, cellularity, and percent of Blasts, Promyelocytes, Basophilis and Eosinophilis, Number of metaphases and additional aberrations for Ph+ and Ph-, for each treatment arm, including Not evaluable or Not Done assessments, will be provided.

## 4.8 SDV sensitivity analysis

In order to assess the impact of patient records-visits with SDV (Source Data Verification) issues, we have performed a sensitivity analysis, excluding specific records involved in SDV issues, for key efficacy and safety outputs. There were 13 patients involved in SDV issues, with 34 visit-records excluded in total.

The following Safety-Efficacy results were repeated:

Study completion-discontinuation, summary of TFR and Re-treatment phase, Molecular response by visit-time window and cumulatively.

Hematology and biochemistry, ECG and Echocardiography summaries. Fasting glucose and Total cholesterol, Vital signs summaries.

Survival and Safety follow-up summaries and Listing of Deaths.

#### 5 Pharmacokinetic evaluations

Not applicable.

## 6 Safety evaluation

Descriptive statistics on AE, laboratory abnormalities, clinically notable ECG, and other safety parameters will be presented as separate outputs. The safety summary tables will include only assessments collected no later than 30 days after study treatment discontinuation.

Safety analysis will be presented per treatment arm and overall during induction/consolidation (between baseline and Month 24 for all patients and between Month 27 and Month 36 for patients randomized in Arm 2). Safety analysis will also be presented per treatment arm and overall during TFR in the subset of patients entering TFR phase and re-treatment phase in the subset of patients entering re-treatment phase.

The safety summary tables will only include events occurring during the treatment periods (see section 2.7.1), while listings will present all assessments (including those occurring during the TFR phase).

#### 6.1 Adverse events

Summary tables will include only TEAEs, i.e. AEs starting or worsening during treatment emergent periods and collected no later than 30 days after study treatment discontinuation. AEs will be coded using the most recent version of the medical dictionary for regulatory activities (MedDRA).

Frequent TEAEs for pre-randomization period, post Randomization (ARM2) and Re-treatment period as well as AEs for TFR period will be summarized in tables. TEAEs, AEs present at 5% or more of the Total group of patients will be classified as Frequent.

The incidence and occurrence of TEAEs (all grades and grades 3 or 4) will be summarized by SOC and PT, as well as the incidence and occurrence of serious TEAEs regardless of their study drug relationship, serious TEAEs suspected to be study drug related, TEAEs leading to study drug discontinuation (only for re-treatment phase), and TEAEs requiring dosage adjustment or temporarily interruption.

Frequent TEAEs and AEs (during TFR), considering events with frequency >=5% for one or more of the treatment Arms, will be presented for pre-randomization induction/consolidation, post randomization consolidation (ARM2), TFR and Re-treatment period. Specifically tables will be created presenting: Overall summary, TEAEs/ AEs by system organ class and preferred term - overall and maximum grade <sup>3</sup>/<sub>4</sub>, Serious Treatment Emergent adverse events regardless of study drug relationship by system organ class and preferred term - overall and maximum grade <sup>3</sup>/<sub>4</sub>. Specific groups of AE of interest will be considered. These are groups of AEs for which there is a specific clinical interest in connection with nilotinib treatment and will be defined through the use of SMQ and PT based on the last version of MedDRA at the time of the analysis. The specific groups to display will be the 4 cardiovascular events (CVEs): CVEs (IHD: Ischemic heart disease), CVEs (PAOD: Peripheral arterial occlusive disease), CVEs (ICE: Ischemic cerebrovascular events) and CVEs (Others). These groups will be defined based on a Novartis project-related document, the "Compound Case Retrieval Strategy" stored in CREDI under path: "Cabinets / CREDI Projects / A / AMN107A / Integrated Medical Safety". The updated version of this document effective at the time of the analysis will be used.

The incidence and occurrence of all grades and grades 3 or 4 of specific TEAEs regardless study drug relationship will be summarized by specific group and PT. These tables on specific AEs will be displayed for the overall FAS, as well as for the 2 following groups of CV risk factors: Very high/High risk; Moderate/Low risk, as well as for each of the CV risk factors separately.

In addition, the time-to-first specific AE (i.e. first occurrence of any of the 4 CVEs defined) will be summarized using Kaplan-Meier estimates and Kaplan-Meier plots will be provided.

Deaths occurring during the treatment emergent period will also be tabulated using SOC and PT (only for re-treatment phase).

All summary tables will be presented separately for pre-randomization induction/consolidation phase (between baseline and Month 24 for all patients), for post-randomization consolidation phase (between Month 27 and Month 36 for patients randomized in Arm 2), and for re-treatment phase. In all incidence summaries, at each level of summarization (specific groups, SOC, and PT), patients will only be counted once regardless of how many times the AE occurred, while in all occurrence summaries, the number of events will be counted.

All AE will also be listed, including those collected during the pre-treatment and post-treatment period (i.e. later than 30 days after study treatment discontinuation). AE occurring outside of the treatment emergent period (during TFR phase) will be flagged and presented separately, since they will not be considered as Treatment Emergent Adverse Events. Listings will detail the verbatim given by the investigator, PT, abbreviated SOC, start date, end date, duration, severity (CTCAE grade), relationship to study drug (not suspected or suspected) and action taken (none, dose adjusted, temporarily interrupted, permanently discontinued, concomitant medication taken, non-drug therapy given, hospitalization/prolonged hospitalization). The AE onset will also be displayed relative (in number of days) to the day of the first dose of study medication. This listing will be repeated for the subsets of serious AEs, AESI and AEs leading to study drug discontinuation.

"TKI withdrawal syndrome" (muscle pain) will be included in the AESI during TFR phase since although related to treatment occurs some days after treatment so it cannot be considered as TEAE.

All deaths will be listed detailing principal cause given by the investigator, PT, date of last dose and date of death. Deaths occurring outside the treatment emergent period will be flagged. The day of last dose and day of death will also be displayed relative to the day of the first dose of study medication. The number of days since last dose (calculated as death day – day of last dose + 1) will also be presented. Also, listing of adverse events leading to study drug discontinuation during re-treatment phase for the subset of FAS entering the re-treatment period will be presented (suggested by SSMC members).

#### 6.2 Laboratory abnormalities

For laboratory tests covered by the CTCAE version 4.03, the laboratory data will be graded accordingly. A Grade 0 will be assigned for all non-missing values not graded as 1 or higher. Grade 5 will not be used.

The following hematological parameters will be graded according to the CTCAE criteria: WBCs, absolute lymphocytes, absolute neutrophils, hemoglobin and platelets.

The following hematological parameters will be classified using normal range: eosinophils, basophils, monocytes, promyelocytes, myelocytes, metamyelocytes and blast.

The following biochemical parameters will be graded according to the CTCAE criteria: bilirubin (total, indirect and direct), aspartate aminotransferase (AST), alanine aminotransferase (ALT), sodium (hyper & hypo), potassium (hyper & hypo), calcium (hyper & hypo), magnesium (hyper & hypo), glucose (hyper & hypo), creatinine, phosphate (or serum phosphorus), lipase, amylase, total cholesterol, triglycerides, alkaline phosphatase (hyper) and albumin (hypo).

The following biochemical parameters will be classified using normal range: HDL, LDL, LDH and HbA1c.

For bi-directional criteria (calcium, glucose, magnesium, potassium and sodium), hyper and hypo abnormalities will be described separately and the value graded in the other direction (e.g. hyper if the parameter of interest is hypo) will be counted as a grade 0.

The following rules will be applied to derive the WBC differential counts when only percentages are available (this is important for neutrophils and lymphocytes, as the CTC grading is based on the absolute counts).

The method to convert the value is as follows: for each patient, the original laboratory value (%) is divided by 100 and multiplied by the WBC count, e.g. for neutrophils (NEU):

NEU count = (WBC count) \* (NEU %value / 100)

In order to derive the corresponding absolute normal range, the rule to be applied depends on the availability of the % range and the absolute range for the differential:

• If the % range is missing and the absolute range is missing, then the pre-defined normal range as reported in the Merck manual (see Novartis business guidance FRM-0015557 - Laboratory value references) will be used.

- If the absolute range is NOT missing (% range is or isn't missing), then the absolute range provided by the site will be used.
- If the % range is NOT missing and the absolute range is missing, then the % normal limits (i.e. lower limit normal (LLN) and upper limit normal (ULN)) are divided by 100 and multiplied by the corresponding normal limits of WBC count, e.g. for NEU:
  - LLN for NEU count = (LLN for WBC count) \* (LLN for NEU % value/ 100)
  - ULN for NEU count = (ULN for WBC count) \* (ULN for NEU % value/ 100)

Shift tables using CTCAE grades will be produced for hematology and biochemistry separately to compare:

- baseline (of induction/consolidation phase) and the worst on-treatment value during post-randomization consolidation phase (see baseline definitions in section 2.4)
- baseline RT and the worst on-treatment value during re-treatment phase (see baseline definitions in section 2.5.3).

Percentages will be calculated using the number of available patients at baseline/baseline RT with corresponding grade and at least one non-missing on-treatment value as the denominator.

Additionally, shift tables between baseline (of induction/consolidation phase) and the worst value during the whole study period (including TFR phase) will be presented.

For laboratory tests where CTCAE grades are not defined, shift tables using the low/normal/high/(low and high) classification will be produced to compare baseline/baseline RT to the worst on-treatment value during respectively induction/consolidation phase and retreatment phase. Percentages will be calculated using the number of available patients at baseline/baseline RT with corresponding classification and at least one non-missing ontreatment value as the denominator.

In addition, descriptive statistics will be provided for all laboratory parameters at each planned visit of the induction/consolidation phase, per treatment arm and overall, and at each planned visit of the re-treatment phase in the subset of FAS entering re-treatment phase.

Listings of hematology and biochemistry laboratory values and normal ranges will be provided, including the sample date/study day, test, SI unit (unit as reported by the site), value, low/high ranges. Grades will also be listed when CTCAE grades are defined.

## 6.3 Vital signs

Vital signs including Height and Weight for Baseline, Body temperature, Sitting pulse and Sitting BP Systolic/Diastolic by visit, will be summarized in tables and will be presented in detailed Listing.

## 6.4 Electrocardiograms (ECGs)

Overall ECG interpretation and details of abnormalities are collected at Screening and selected visits. The ECG QTcF result (msec) at each visit will be categorized ( $\leq$ 450, >450 - $\leq$ 480, >480 -  $\leq$ 500, >500 and missing). Shift tables will display the categorized ECG QTcF result at baseline/baseline RT compared to the worst on-treatment value during respectively induction/consolidation phase and re-treatment phase.

A shift table displaying the baseline categorized ECG QTcF result compared with the worst post-baseline categorized result will be produced. Percentages will be calculated using the number of patients with that categorized result at baseline as the denominator.

The number of patients recording notable ECG QTcF increases (Increase from baseline > 30/ Increase from baseline > 60) from baseline/baseline RT at least once during the trial will also be presented. Percentages will be calculated using the number of patients with both baseline/baseline RT and post baseline/baseline RT evaluations.

A listing will be provided including the date of ECG, QTcF interval, and whether there is a clinically significant abnormality

## 6.5 Echocardiography (cardiac imaging)

As per protocol, echocardiography is performed at screening and may be repeated at the investigator's discretion if there are signs or symptoms of cardiotoxicity.

Baseline LVEF data will be descriptively analyzed, together with the overall interpretation (normal, clinically insignificant abnormality, clinically significant abnormality). A shift table displaying the baseline overall interpretation compared with the worst post-baseline overall interpretation will be produced. Percentages will be calculated using the number of patients with that overall interpretation at baseline as the denominator.

## 6.6 Survival Follow-up

Survival follow-up records will be summarized in a table by FU visit, presenting frequency as number and percentage of alive patients, Cases of stem cell transplantation, Progression of disease to AP/BP, administration of TKI treatment and drug category (Nilotinib, Imatinib, Other) if yes.

Time window for Survival follow-up defined in section 2.5.1.

A listing will be provided presenting for each visit: subject status (alive yes /no), if no date of death and principal cause of death along with specific details in case of other cause. If subject alive or lost to follow-up last date of contact will be presented. Information regarding stem cell transplantation, Progression of disease to AP/BP, administration of TKI treatment and drug category (Nilotinib, Imatinib, Other) if yes, along with specific details for treatment in case of other than standard categories.

## 6.7 Safety Follow-up

Safety follow-up information will be summarized in a table of frequency as number and percentage, including: type of follow-up (clinical visit, telephone call), as well as if Medical intervention was considered necessary.

A listing will be provided including all relevant information collected in the CRF:

If follow-up happened, if no reason for no safety follow-up, if yes, type of follow-up (clinical visit, telephone call), along with the respective date. If Medical intervention was considered necessary and date of Medical intervention.

## 6.8 LSC sub-study analysis

Apart from selected parts of the main study analysis that will be repeated for patients participating in the LSC sub-study in addition will be presented:

Descriptive Statistics for Baseline, Months 24, 36, EOP TFR as well as for change from baseline for:

- CD34 cells as Total percentage.
- CD34+/CD38+ cells Percentage from total CD34+ cells.
- Descriptive Statistics for number of events sorted in CD34+/CD38+ cells

Then proportion and descriptive statistics tables for patients with presence of Ph+ LSC in bone marrow, in terms of in CD34+/CD38+, CD34+/CD38-, Immunophenotypically aberrant CD34+ and Immunophenotypically aberrant CD34 negative cells as:

- Ph+ by HIS status,
- Descriptive statistics of Ph+ in CD34+/CD38+ cells
- BCR-ABL by RT-PCR status, in CD34+/CD38+ cells

#### Specifically:

- Percentage from total CD34+ cells, CD34+/CD38+ cells.
- Percentage from total CD34+ cells, CD34+/CD38- cells.
- Percentage from total CD34+ cells.
- Percentage from total CD34+ cells.
- Percentage of Ph+ cells, CD34+/CD38+ cells.
- Percentage of Ph+ cells, CD34+/CD38- cells.
- Percentage of Ph+ cells, Immunophenotypically aberrant CD34+ cells.
- Percentage of Ph+ cells, Immunophenotypically aberrant CD34 negative cells.
- Total Percentage of CD34+ cells.

Frequency and descriptive statistics tables will be created for the above endpoints, along with Listings presenting individual data.

For the 24/36 month data analysis for the Leukemic Stem Cell sub-study of the CAMN107AIC05 clinical trial, additional analysis will be performed for publication purposes. Prior Imatinib exposure before screening (<5 vs >=5 years), Major Molecular Response (MMR Yes vs No), Age (<65 vs >=60 years) and Sokal score (Low, Intermediate, High risk) by LSC category at Baseline, will be presented for Not Randomized and Randomized patients in a summary table.

Tables summarizing descriptive statistics of LSC cells for Baseline, Month 24 as well as the change from Baseline to Month 24, will be presented for Arm1, Arm2, Not Randomized, Randomized (Arm1 and Arm2) and Total (Randomized and Not Randomized), for LSC detected subjects.

A table presenting number and percentage of subjects using separate columns for Arm1, Arm2, Not Randomized, Randomized (Arm1 and Arm2) and Total (Randomized and Not Randomized), at Baseline, Month 24, Month 36 (for Arm 2 subjects only) and EOP TFR will be created.

In addition, individual figures for HIS and PCR detected patients, presenting number of sorted events for each patient by visit (Baseline, Month 24, Month 36 for ARM2 patients only and EOP TFR), will be provided. Separate figures for each one of the 4 basic cell categories will be presented:

- CD34+/CD38+
- CD34+ / CD38-
- Immunophenotypically aberrant CD34+
- Immunophenotypically aberrant CD34-

Summary figures will be created, presenting number and percentage of patients with positive result by HIS and PCR by visit (Baseline, Month 24, Month 36 for ARM2 patients only and EOP TFR) for :

- CD34+/CD38+
- CD34+/CD38-
- Immunophenotypically aberrant CD34+
- Immunophenotypically aberrant CD34-

Number of patients with detectable LSC – LSC sub study for LSCFAS will be presented by bar diagram for publication purpose.

# 7 Other topics

No other topics will be studied.

# 8 Sample size calculation

According to the protocol amendment 2, it is expected that approximately 565 patients from approximately 300 centers will be recruited into this study.

This sample size calculation has been based on an estimation of the difference in the percentage of patients relapsing during the 12-month TFR phase of the study between the two treatment arms. Further details are given in the study protocol.

#### 9 References

Protocol AMN107AIC05, version 04 (including Amendment 4); 01 Jun 2016.

Common Terminology Criteria for Adverse Events (CTCAE), version 4.03, US Department of Health and Human Services, National Institutes of Health, National Cancer Institute, NIH Publication No. 09-5410, published on May 28, 2009 (v4.03: June 14, 2010)

http://evs.nci.nih.gov/ftp1/CTCAE/CTCAE 4.03 2010-06-14 QuickReference 5x7.pdf

Merck Manual of Therapeutics, Normal Laboratory Values; FRM-0015557 v 3.0.

European Guidelines on cardiovascular disease prevention in clinical practice (version 2012). European Heart Journal (2012) 33, 1635–1701



# Clinical Development & Medical Affairs

# AMN107 (Nilotinib, Tasigna®)

Study Number: CAMN107AIC05/NCT01743989

A prospective, randomized, open-label, two-arm Phase III study to evaluate treatment-free remission (TFR) rate in patients with Philadelphia chromosome-positive CML after two different durations of consolidation treatment with nilotinib 300 mg BID

#### RAP Module 7.1- CSR deliverables

Authors: Statistician

, Novartis study statistician

Document type: RAP Documentation

Document status: Addendum 2

Release date: 06-May-2021

Number of pages: 425

Property of Novartis
May not be used, divulged, published or otherwise disclosed without the consent of Novartis

# **Document History – Changes compared to previous version of RAP module 7.1**

| Version | <br>Date | Changes |
|---|---|---|
| | | Changes |
| 1.0 | 08-Jan-2020 | First Draft |
| 1.1 | 10-Feb-2020 | Updated version, added LSC substudy ouputs |
| 1.2 | 05-Mar-2020 | Revised version |
| 1.3 | 20-Mar-2020 | Updated version after tema review |
| 1.4 | 23-Apr-2020 | Updated tables with PPS outputs, added LSC extra analysis |
| 1.5 | 17-Jun-2020 | Updated according to DR1 findings |
| 1.6 | 31-Aug-2020 | Updated according to DR2 findings |
| 1.7 | 22-Sep-2020 | Updated according to Final Run requirements |
| 1.8 | 06-Oct-2020 | Added SSMC requested outputs |
| Pre-Final | 07-Oct-2020 | Finalize document |
| Final | 09-Oct-2020 | Minor cosmetics update and final version for CSR |
| Addendum | 18-Jan-2021 | Sensitivity analysis, repeat key outputs excluding SDV(not done) involved visits, footnotes updated for populations as per module 3, Updated KM TLFs for progression to AP/BC (eCRF captured variable) for PFS and TFS. In text tables footnotes are shortned in outputs. Table numbers are updated for following: T14.2-4.2.1.1 to T14.2-4.2.11, T14.3-1.1.2.1 to T14.3-1.1.21, T14.3-1.1.2.2 to T14.3-1.1.22, Figure numbers are updated for following: F14.2-2.3.1.1 to F14.2-2.3.11, F14.2-2.5.1.1 to F14.2-2.5.11 |
| | | Cut off date in TLFs footnotes replaced by DBL date Minor updates in title and footnote as per CSR final run review comments. |
| Addendum<br>V1.1 | 29-Jan-2021 | Excluding Safety SDV analysis outputs as they were not affected by the SDV record exclusion of specific visits, since they are based on Start and Stop dates independently of standard study visits. Tables 14.3-1.1.4 and 14.3-2.4, 14.3-3.4, 14.3-4.5 and 14.3-4.6 for Duration of exposure, Relative dose intension, Dose reduction, Concomitant medication during TFR and Re-treatment. Tables 14.3.1-1.5, 14.3.1-3.3.3, 14.3.1-4.3.3, 14.3.1-4.4.3 14.3.1-4.8.3, 14.3.1-5.3.3, 14.3.1-6.3.3, 14.3.1-6.6.3, 14.3.1-6.7.3, 14.3.1-7.3.3, 14.3.1-7.4.3, 14.3.1-7.8.3 for AEs and TEAEs. Table 14.3.1-9.4 for On treatment deaths. Tables 14.3.1-10.3.3, 14.3.1-10.4.3, 14.3.1-10.7, 14.3.1-10.8 and 14.3.1-11.3 for CVEs. Table 14.3.1-12.2 for Medical History. Figures 14.3.1-1.5 and 1.6 for Time to CVE. |
| Addendum<br>V1.2 | 09-Mar-2021 | Adding footnote for patient # in Tables: 10-2,14.1-2.1, 14.1-2.5, 14.1-2.6, 14.1-2.6.1, 12-1, 14.3.1-1.1,14.3.1-2.1, 14.3.1-3.1.1, 14.3.1-3.1.2,14.3.1-3.5.1, 14.3.1-4.1.1, 14.3.1-4.1.2, 14.3.1-4.6.1, 14.3.1-4.6.2 12-17, 14.3.1-5.1.1, 14.3.1-5.1.2, 14.3.1-6.1.1, 14.3.1-6.1.2 Listings: 14.3.2-2.2, 16.2.7-1.1, 16.2.7-2.2, 16.2.1-1.1, 16.2.1-1.2, 16.2.5-1.1 |

| Version | Date | Changes |
|---|---|---|
| | | Adding footnote for patient in tables: 12-1, 12-9 14.3.1-1.1, 14.3.1-1.2, 14.3.1-2.1, 14.3.1-3.1.1, 14.3.1-3.1.2, 14.3.1-4.1.1, 14.3.1-4.1.2, 14.3.1-4.6.1, 14.3.1-4.6.2, 14.3.1-6.1.1, 14.3.1-6.1.2 Listings: 16.2.7-1.1, 16.2.7-2.1 |
| Addendum<br>V1.3 | 20-Apr-2021 | Adding footnote for patient # in tables: 12-1, 12-9, 12-17 14.3.1-1.1, 14.3.1-1.2, 14.3.1-2.1, 14.3.1-3.1.1, 14.3.1-3.1.2, 14.3.1-4.1.1, 14.3.1-4.1.2, 14.3.1-4.6.1, 14.3.1-4.6.2, 14.3.1-5.1.1, 14.3.1-5.1.2, 14.3.1-6.1.1, 14.3.1-6.1.2 Lietings: 14.3.2.2.2, 16.3.7.1, 16.3.7.2.1, 16.3.7.2.2 |
| | | Listings: 14.3.2-2.2, 16.2.7-1.1, 16.2.7-2.1, 16.2.7-2.2 Adding footnote for patient # in tables: 14.1-2.2, 14.1-2.5, 14.1-2.6 and 14.1-2.6.1 |
| Addendum<br>V1.4 | 06-May-2021 | Adding Listing 16.1.7-1.1 Randomization schemes on Randomized patients |
| Addendum 2 | 06-May-2021 | Final version |


| Table 12-1 Overall summary of treatment-emergent adverse events occurring during pre-randomization Induction/consolidation phase – Full Analysis Set | 2 |
|---|---|
| Table 12-2 Overall summary of treatment-emergent adverse events occurring during post-randomization consolidation phase (ARM 2) – Subset of Full Analysis Set randomized to Arm 2 | 3 |
| Table 12-3 Overall summary of treatment-emergent adverse events occurring during re-treatment phase – Subset of Full Analysis Set entering the re-treatment phase | 4 |
| Table 12-4 Overall summary of adverse events occurring during TFR phase – Subset of Full Analysis Set entering the TFR phase | 5 |
| Table 12-5 Overall summary of frequent [1] treatment-emergent adverse events occurring during pre-randomization Induction/consolidation phase – Full Analysis Set | 6 |
| Table 12-6 Overall summary of frequent [1] treatment-emergent adverse events occurring during post-randomization Consolidation phase (ARM 2) – Subset of Full Analysis Set randomized to Arm 2 | 6 |
| Table 12-7 Overall summary of frequent [1] treatment-emergent adverse events occurring during re-treatment phase — Subset of Full Analysis Set entering the re-treatment phase — 120 | 6 |
| Table 12-8 Overall summary of frequent [1] adverse events occurring during TFR phase – Subset of Full Analysis Set entering the TFR phase | 6 |
| Table 12-9 Serious treatment-emergent adverse events incidence, regardless of study drug relationship, by system organ class and preferred term during prerandomization Induction/consolidation phase – overall and maximum grade 3/4 –Full Analysis Set | 7 |
| Table 12-10 Serious treatment-emergent adverse events incidence, regardless of study drug relationship, by system organ class and preferred term during post-randomization consolidation phase (ARM 2) – overall and maximum grade 3/4 – Subset of Full Analysis Set randomized to Arm 2 | 8 |
| Table 12-11 Serious treatment-emergent adverse events incidence, regardless of study drug relationship, by system organ class and preferred term during retreatment phase — overall and maximum grade 3/4 — Subset of Full Analysis Set entering the re-treatment phase | 8 |
| Table 12-12 Serious adverse events incidence, regardless of study drug relationship, by system organ class and preferred term during TFR phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the TFR phase 120 | 8 |
| Table 12-13 Treatment-emergent adverse events of interest incidence, regardless of study drug relationship, by specific group and preferred term during Prerandomization Induction/consolidation phase –by treatment arm, overall and maximum grade 3/4 – Full Analysis Set | 9 |
| Table 12-14 Treatment-emergent adverse events of interest incidence by specific group and preferred term during post-randomization Consolidation phase (ARM 2) – overall and maximum grade 3/4 – Subset of Full Analysis Set | 0 |

| Table 12-15 Treatment-emergent adverse events of interest incidence by specific group and preferred term during re-treatment phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the re-treatment phase | .131 |
|---|---|
| Table 12-16 Adverse events of interest incidence by specific group and preferred term during TFR phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the TFR phase | 131 |
| Table 12-17 Treatment-emergent adverse events incidence leading to study drug discontinuation by system organ class and preferred term during prerandomization Induction/Consolidation phase – overall and maximum grade 3/4 –Full Analysis Set | .132 |
| Table 12-18 Treatment-emergent adverse events incidence leading to study drug discontinuation by system organ class and preferred term during post-randomizationphase (ARM 2) – overall and maximum grade 3/4 – Subset of Full Analysis Set randomized to Arm 2 | .133 |
| Table 12-19 On treatment deaths, by system organ class and preferred term during pre-randomization Induction/Consolidation phase - Safety Set | 133 |
| Table 12-20 On treatment deaths, by system organ class and preferred term during post-randomization consolidation phase (ARM 2) – Subset of Safety Set randomized to Arm 2 | 134 |
| Table 12-21 On treatment deaths, by system organ class and preferred term during re-treatment phase – Subset of Safety Set entering the re-treatment phase | .134 |
| Listing 12-1 Listing of deaths – Full Analysis Set | .135 |
| Figure 11-1 Primary endpoint, Bar plot MR4.0 at 12 months of TFR phase —Subset of Full Analysis Set entering the TFR phase | 136 |
| Figure 11-2 Kaplan-Meier analysis of treatment-free survival during the TFR phase -Subset of Full Analysis Set entering the TFR phase | 137 |
| 3.2 Shells and specifications for Sections 14 and 16 of the CSR | .138 |
| Section 14 – tables, figures and graphs referred to but not included in the text | |
| Section 14.1 – Demographic data | 138 |
| Table 14.1-1.1 Enrollment by country and center – All patients | |
| Table 14.1-1.2 Randomization by country and center – Randomized patients | |
| Table 14.1-1.3 Patient disposition (Screening failures), All patients | .141 |
| Table 14.1-2.1 Patient disposition during Induction/Consolidation phase and post-Randomization Consolidation phase -Enrolled patients | |
| Table 14.1-2.2 Patient disposition in each randomized arm – Full Analysis Set | |
| Table 14.1-2.2.1 Patient disposition – Enrolled patients in LSC substudy | |
| Table 14.1-2.3 Analysis sets –All patients | |
| Table 14.1-2.4 Not Randomized patients - Enrolled patients | |
| Table 14.1-2.5 Patient disposition, Overall and by year-phase -Enrolled patients | |
| Table 14.1-2.6 Patients discontinued and reason for discontinuation – Full Analysis | |
| Set | .134 |
| Table 14.1-2.6.1 Patients discontinued and reason for discontinuation, SDV sensitivity – Full Analysis Set | .156 |

| Table 14.1-2.7 Summary of TFR phase – Full Analysis Set | .157 |
|---|---|
| Table 14.1-2.7.1 Summary of TFR phase, SDV sensitivity – Full Analysis Set | |
| Table 14.1-2.8 Summary of re-treatment phase – Full Analysis Set | .159 |
| Table 14.1-2.8.1 Summary of re-treatment phase, SDV sensitivity – Full Analysis Set | .160 |
| Table 14.1-2.9 Summary of patients with relapse during the TFR phase but no entering re-treatment phase —Subset of Full Analysis Set entering the TFR phase | 161 |
| Table 14.1-3.1 Demographic and characteristics at baseline– Full Analysis Set | |
| Table 14.1-3.1.1 Demographic and characteristics at baseline– LSC sub-study Full | |
| Analysis Set | |
| Table 14.1-4.1 Disease history – Full Analysis Set. | |
| Table 14.1-4.1.1 Disease history – LSC sub-study Full Analysis Set. | |
| Table 14.1-5.1 History of prior Imatinib therapy – Full Analysis Set | |
| Table 14.1-5.1.1 History of prior Imatinib therapy – LSC sub-study Full Analysis Set. | .1/2 |
| Table 14.1-5.2 Prior antineoplastic therapy, other than Imatinib, by ATC class and preferred term - Full Analysis Set | .173 |
| Table 14.1-6.1 Cardiovascular risk factors at baseline – Full Analysis Set | |
| Table 14.1-6.2 Cardiovascular risk factors (based on medical history, laboratory | |
| values and vital signs at baseline) – Full Analysis Set | .175 |
| Section 14.2 – Efficacy and other non-safety data (e.g. PK, PK/PD, Health Econ., QoL) | .177 |
| Figure 14.2-1.1 Box-plot of BCR-ABL ratio (IS) during pre-randomization Induction/Consolidation phase – Full Analysis Set | .178 |
| Figure 14.2-1.2 Box-plot of BCR-ABL ratio (IS) during post-randomization<br>Consolidation phase (ARM 2) – Subset of Full Analysis Set randomized to<br>ARM 2 | .179 |
| Figure 14.2-1.3 Box-plot of BCR-ABL ratio (IS) during TFR phase – Subset of Full Analysis Set entered TFR | .179 |
| Figure 14.2-1.4 Box-plot of BCR-ABL ratio (IS) during re-treatment phase – Subset of Full Analysis Set entered re-treatment | .179 |
| Figure 14.2-1.5 Box-plot of BCR-ABL ratio (IS) during TFR phase – , SDV sensitivity Subset of Full Analysis Set entered TFR | .180 |
| Figure 14.2-1.6 Box-plot of BCR-ABL ratio (IS) during re-treatment phase, SDV sensitivity –Subset of Full Analysis Set entered re-treatment | .180 |
| Figure 14.2-2.1.1 Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase - Full Analysis Set | .181 |
| Figure 14.2-2.1.2 Raw cumulative incidence of MMR during post-randomization Consolidation phase (ARM 2) - Subset of Full Analysis Set randomized to ARM 2 | .181 |
| Figure 14.2-2.2.1 Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase by halving time of BCR-ABL (IS) ratio - Full Analysis Set | 182 |

| Figure | 14.2-2.2.2 Raw cumulative incidence of MMR during post-randomization Consolidation phase (ARM 2) by halving time of BCR-ABL (IS) ratio - Subset of Full Analysis Set randomized to ARM 2 | 182 |
|---|---|---|
| Figure | 14.2-2.3.1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase – Full Analysis Set | 183 |
| Figure | 14.2-2.3.2 Raw cumulative incidence of MR 4.0 during post-randomization Consolidation phase (ARM 2) - Subset of Full Analysis Set randomized to ARM 2 | 183 |
| Figure | 14.2-2.3.11 Raw cumulative incidence of MR 4.0, Randomized vs Not Randomized, during pre-randomization Induction/Consolidation phase - Full Analysis Set | 184 |
| Figure | 14.2-2.4.1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase by halving time of BCR-ABL (IS) ratio - Full Analysis Set | 184 |
| Figure | 14.2-2.4.2 Raw cumulative incidence of MR 4.0 during post-randomization Consolidation phase (ARM 2) by halving time of BCR-ABL (IS) ratio - Subset of Full Analysis Set randomized to ARM 2 | 185 |
| Figure | 14.2-2.5.1 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase - Full Analysis Set | 185 |
| Figure | 14.2-2.5.11 Raw cumulative incidence of MR 4.5, Randomized vs Not Randomized, during pre-randomization Induction/Consolidation phase-Full Analysis Set | 185 |
| Figure | 14.2-2.5.2 Raw cumulative incidence of MR 4.5 during post-randomization Consolidation phase (ARM 2) - Subset of Full Analysis Set randomized to ARM 2 | 185 |
| Figure | 14.2-2.6.1 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase by halving time of BCR-ABL (IS) ratio - Full Analysis Set | 185 |
| Figure | 14.2-2.6.2 Raw cumulative incidence of MR 4.5 during post-randomization Consolidation phase (ARM 2) by halving time of BCR-ABL (IS) ratio - Subset of Full Analysis Set randomized to ARM 2 | 186 |
| Figure | 14.2-2.7.1 Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase - Full Analysis Set patients not reaching MMR at baseline | 186 |
| Figure | 14.2-2.8.1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase - Full Analysis Set patients not reaching MR 4.0 at baseline | |
| Figure | 14.2-2.9.1 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase - Full Analysis Set patients not reaching MR 4.5 at baseline | |
| Figure | 14.2-2.9.2 Raw cumulative incidence of MR 4.5 during post-randomization Induction/Consolidation phase (ARM 2)- Subset of Full Analysis Set patients not reaching MR 4.5 at baseline, randomized to ARM 2 | 186 |
| Figure | 14.2-2.10.1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase by BCR-ABL(IS) ratio at baseline - Full Analysis Set | 187 |

| Figure | 14.2-2.10.2 Raw cumulative incidence of MR 4.0 during post-randomization Consolidation phase (ARM 2) by BCR-ABL(IS) ratio at baseline - Subset of Full Analysis Set randomized to ARM 2 | 187 |
|---|---|---|
| Figure | 14.2-2.11.1 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase by BCR-ABL(IS) ratio at baseline - Full Analysis Set | 188 |
| Figure | 14.2-2.11.2 Raw cumulative incidence of MR 4.5 during post-randomization Consolidation phase (ARM 2) by BCR-ABL(IS) ratio at baseline - Subset of Full Analysis Set randomized to ARM 2 | 188 |
| Figure | 14.2-2.12.1 Box-plot of BCR-ABL ratio (IS) during pre-randomization Induction/Consolidation phase, excluding outliers (BCR-ABL (IS) ratio>10 - Full Analysis Set | 189 |
| Figure | 14.2-2.12.2 Box-plot of BCR-ABL ratio (IS) over post-randomization Consolidation phase (ARM 2), excluding outliers (BCR-ABL (IS) ratio>10 - Subset of Full Analysis Set randomized to ARM 2 | 189 |
| Figure | 14.2-13.1 Raw cumulative incidence of loss of MMR during TFR – Subset of Full Analysis Set entering the TFR phase | 191 |
| Figure | 14.2-13.2 Raw cumulative incidence of MMR during re-treatment phase – Subset of Full Analysis Set entering the re-treatment phase | 191 |
| Figure | 14.2-13.3 Raw cumulative incidence of loss of MMR during TFR, SDV sensitivity – Subset of Full Analysis Set entering the TFR phase | 192 |
| Figure | 14.2-13.4 Raw cumulative incidence of MMR during re-treatment phase, SDV sensitivity – Subset of Full Analysis Set entering the re-treatment phase1 | 192 |
| Figure | 14.2-14.1 Raw cumulative incidence of loss of MR4.0 during TFR phase – Subset of Full Analysis Set entering the TFR phase | 192 |
| Figure | 14.2-14.2 Raw cumulative incidence of MR4.0 during re-treatment phase – Subset of Full Analysis Set entering the re-treatment phase | 192 |
| Figure | 14.2-14.3 Raw cumulative incidence of loss of MR4.0 during TFR phase, SDV sensitivity –Subset of Full Analysis Set entering the TFR phase | 193 |
| Figure | 14.2-14.4 Raw cumulative incidence of MR4.0 during re-treatment phase, SDV sensitivity – Subset of Full Analysis Set entering the re-treatment phase1 | 193 |
| Figure | 14.2-15.1 Raw cumulative incidence of loss of MR4.5 during TFR phase – Subset of Full Analysis Set entering the TFR phase with MR4.5 | 193 |
| Figure | 14.2-15.2 Raw cumulative incidence of MR4.5 during re-treatment phase – Subset of Full Analysis Set entering the re-treatment phase | |
| Figure | 14.2-15.3 Raw cumulative incidence of loss of MR4.5 during TFR phase, SDV sensitivity – Subset of Full Analysis Set entering the TFR phase with MR4.5 | |
| Figure | 14.2-15.4 Raw cumulative incidence of MR4.5 during re-treatment phase, SDV sensitivity – Subset of Full Analysis Set entering the re-treatment phase1 | 194 |
| Figure | 14.2-16 Bar plot MR4.0 at 12 months of TFR phase —Subset of Full Analysis Set entering the TFR phase ———————————————————————————————————— | |
| Figure | 14.2-16.2 Bar plot MR4.0 at month 12 TFR phase, SDV sensitivity –Subset of Full Analysis Set entering the TFR phase | |

| Figure 14.2-17.1 Kaplan-Meier analysis of progression-free survival during the TFR phase –Subset of Full Analysis Set entering the TFR phase | .196 |
|---|---|
| Figure 14.2-17.2 Kaplan-Meier analysis of treatment-free survival during the TFR phase –Subset of Full Analysis Set entering the TFR phase | .196 |
| Figure 14.2-17.3 Kaplan-Meier analysis of progression-free survival during the TFR phase, SDV sensitivity –Subset of Full Analysis Set entering the TFR phase | .197 |
| Figure 14.2-17.4 Kaplan-Meier analysis of treatment-free survival during the TFR phase, SDV sensitivity –Subset of Full Analysis Set entering the TFR phase | .197 |
| Figure 14.2-18.1 Kaplan-Meier analysis of reachievement of MMR, after loss of response in TFR –Subset of Full Analysis Set entering the re-treatment phase. | .197 |
| Figure 14.2-18.2 Kaplan-Meier analysis of reachievement of MR4.0, after loss of response in TFR – Subset of Full Analysis Set entering the re-treatment phase | .197 |
| Figure 14.2-18.3 Kaplan-Meier analysis of reachievement of MMR, after loss of response in TFR, SDV sensitivity –Subset of Full Analysis Set entering the re-treatment phase | .198 |
| Figure 14.2-18.4 Kaplan-Meier analysis of reachievement of MR4.0, after loss of response in TFR, SDV sensitivity – Subset of Full Analysis Set entering the re-treatment phase | .198 |
| Table 14.2-1.1 Description of BCR-ABL (IS) ratio at Month 3 and halving time of BCR-ABL (IS) ratio subgroups – Full Analysis Set | .199 |
| Table 14.2-2.1.1 Molecular response MR4.0 at 12 months of TFR–Subset of Full Analysis Set entering the TFR phase | .200 |
| Table 14.2-2.1.2 Molecular response MR4.0 at 12 months of TFR–Subset of Per Protocol Analysis Set entering the TFR phase | .200 |
| Table 14.2-2.1.3 Molecular response MR4.0 at 12 months of TFR-Full Analysis Set. | .201 |
| Table 14.2-2.1.4 Molecular response MR4.0 at 12 months of TFR–Per Protocol Analysis Set | .201 |
| Table 14.2-2.1.5 Molecular response MR4.0 at 12 months of TFR—Subset of Full Analysis Set entering the TFR phase with MR4.0 achieved up to month 3 of pre-randomization Induction/Consolidation phase | .202 |
| Table 14.2-2.1.6 Molecular response MR4.0 at 12 months of TFR—Subset of Full Analysis Set entering the TFR phase with MR4.5 achieved up to month 3 of pre-randomization Induction/Consolidation phase | .202 |
| Table 14.2-2.1.7 Molecular response MR4.0 at 12 months of TFR, SDV sensitivity – Subset of Full Analysis Set entering the TFR phase | |
| Table 14.2-2.1.8 Molecular response MR4.0 at 12 months of TFR, SDV sensitivity – Subset of Per Protocol Analysis Set entering the TFR phase | |
| Table 14.2-2.1.9 Molecular response MR4.0 at 12 months of TFR, SDV sensitivity – Full Analysis Set | |
| Table 14.2-2.1.10 Molecular response MR4.0 at 12 months of TFR, SDV sensitivity —Per Protocol Analysis Set | .203 |
| Table 14.2-2.2.1 Kaplan-Meier analysis of treatment-free survival during the TFR phase – Subset of Full Analysis Set entering the TFR phase | .204 |

| Table 14.2-2.2.2 Kaplan-Meier analysis of treatment-free survival during the TFR phase – Subset of Per Protocol Analysis Set entering the TFR phase | 205 |
|---|---|
| Table 14.2-2.2.3 Kaplan-Meier analysis of treatment-free survival during the TFR phase, SDV sensitivity – Subset of Full Analysis Set entering the TFR phase | 205 |
| Table 14.2-2.2.4 Kaplan-Meier analysis of treatment-free survival during the TFR phase, SDV sensitivity – Subset of Per Protocol Analysis Set entering the TFR phase | 205 |
| Table 14.2-2.3 Kaplan-Meier analysis of overall survival from Randomization— Randomized Set | 206 |
| Table 14.2-2.4 Kaplan-Meier analysis of progression-free survival during the TFR phase — Subset of Full Analysis Set entering the TFR phase | 207 |
| Table 14.2-2.5 Kaplan-Meier analysis of overall survival from Randomization, SDV sensitivity –Randomized Set | 208 |
| Table 14.2-2.6 Kaplan-Meier analysis of progression-free survival during the TFR phase, SDV sensitivity — Subset of Full Analysis Set entering the TFR phase. | 208 |
| Table 14.2-3.1 Major molecular response during pre-randomization Induction/Consolidation phase –Full Analysis Set | 209 |
| Table 14.2-3.1.1 Major molecular response during pre-randomization<br>Induction/Consolidation phase – LSC sub-study Full Analysis Set | 210 |
| Table 14.2-3.2 Major molecular response during post-randomization consolidation phase (ARM 2)— Subset of Full Analysis Set randomized to Arm 2 | 211 |
| Table 14.2-3.2.1 Major molecular response during post-randomization consolidation phase (ARM 2) – LSC sub-study Full Analysis Set randomized to Arm 2 | 211 |
| Table 14.2-3.3 Major molecular response during TFR phase —Subset of Full Analysis Set patients entered TFR phase | 212 |
| Table 14.2-3.4 Major molecular response during re-treatment phase—Subset of Full Analysis Set patients entered re- treatment phase | 213 |
| Table 14.2-3.5 Major molecular response during TFR phase –Subset of Full Analysis Set patients entered TFR phase with MR4.0 achieved up to month 3 of prerandomization Induction/Consolidation phase | 214 |
| Table 14.2-3.6 Major molecular response during TFR phase –Subset of Full Analysis Set patients entered TFR phase with MR4.5 achieved up to month 3 of prerandomization Induction/Consolidation phase | 214 |
| Table 14.2-3.7 Major molecular response during TFR phase, SDV sensitivity – Subset of Full Analysis Set patients entered TFR phase | 214 |
| Table 14.2-3.8 Major molecular response during re-treatment phase, SDV sensitivity —Subset of Full Analysis Set patients entered re- treatment phase | 214 |
| Table 14.2-4.1 Molecular response 4.0 during pre-randomization<br>Induction/Consolidation phase – Full Analysis Set | 215 |
| Table 14.2-4.1.1 Molecular response 4.0 during pre-randomization<br>Induction/Consolidation phase – LSC sub-study Full Analysis Set | 215 |
| Table 14.2-4.2.1 Molecular response 4.0 during post-randomization consolidation phase (ARM 2) – Subset of Full Analysis Set randomized to Arm 2 | 215 |

| Table 14.2-4.2.2 Molecular response 4.0 during post-randomization consolidation phase (ARM 2) – Subset of Per Protocol randomized to Arm 2 | 215 |
|---|---|
| Table 14.2-4.2.11 Molecular response 4.0 during post-randomization consolidation phase (ARM 2) – Subset of LSC sub-study Full Analysis Set randomized to Arm 2 | 215 |
| Table 14.2-4.3.1 Molecular response 4.0 during TFR phase – Subset of Full Analysis Set entering the TFR phase | |
| Table 14.2-4.3.2 Molecular response 4.0 during TFR phase – Subset of Per Protocol Analysis Set entering the TFR phase | 216 |
| Table 14.2-4.3.3 Molecular response 4.0 during TFR phase , SDV sensitivity – Subset of Full Analysis Set entering the TFR phase | 216 |
| Table 14.2-4.4 Molecular response 4.0 during re-treatment phase – Subset of Full Analysis Set entering the re-treatment phase | 217 |
| Table 14.2-4.5 Molecular response 4.0 during TFR phase – Subset of Full Analysis Set entering the TFR phase with MR4.0 achieved up to month 3 of prerandomization Induction/Consolidation phase | 217 |
| Table 14.2-4.6 Molecular response 4.0 during TFR phase – Subset of Full Analysis Set entering the TFR phase with MR4.5 achieved up to month 3 of prerandomization Induction/Consolidation phase | 217 |
| Table 14.2-4.7 Molecular response 4.0 during re-treatment phase, SDV sensitivity – Subset of Full Analysis Set entering the re-treatment phase | 217 |
| Table 14.2-5.1 Molecular response 4.5 during pre-randomization Induction/Consolidation—Full Analysis Set | 218 |
| Table 14.2-5.1.1 Molecular response 4.5 during pre-randomization Induction/Consolidation— LSC sub-study Full Analysis Set | 218 |
| Table 14.2-5.2 Molecular response 4.5 during post-randomization consolidation phase (ARM 2) – Subset of Full Analysis Set randomized to Arm 2 | 218 |
| Table 14.2-5.2.1 Molecular response 4.5 during post-randomization consolidation phase (ARM 2) – Subset of LSC sub-study Full Analysis Set randomized to Arm 2 | 218 |
| Table 14.2-5.3 Molecular response 4.5 during TFR phase – Subset of Full Analysis Set entering the TFR phase | 218 |
| Table 14.2-5.4 Molecular response 4.5 during re-treatment phase – Subset of Full Analysis Set entering the re-treatment phase | 218 |
| Table 14.2-5.5 Molecular response 4.5 during TFR phase – Subset of Full Analysis Set entering the TFR phase with MR4.0 achieved up to month 3 of prerandomization Induction/Consolidation phase | 219 |
| Table 14.2-5.6 Molecular response 4.5 during TFR phase – Subset of Full Analysis Set entering the TFR phase with MR4.5 achieved up to month 3 of prerandomization Induction/Consolidation phase | 219 |
| Table 14.2-5.7 Molecular response 4.5 during TFR phase, SDV sensitivity – Subset of Full Analysis Set entering the TFR phase | 219 |
| Table 14.2-5.8 Molecular response 4.5 during re-treatment phase, SDV sensitivity – Subset of Full Analysis Set entering the re-treatment phase | 219 |

| Table 14.2-6.1 Raw cumulative incidence MMR during pre-randomization Induction/Consolidation phase – Full Analysis Set |
|---|
| Table 14.2-6.1.1 Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase – LSC sub-study Full Analysis Set221 |
| Table 14.2-6.2 Raw cumulative incidence MMR during post-randomization Consolidation phase (ARM 2) - Subset of Full Analysis Set patients randomized to ARM 2 |
| Table 14.2-6.2.1 Raw cumulative incidence MMR during post-randomization Consolidation phase (ARM 2) - Subset of LSC sub-study Fulls Anslysis Set randomized to ARM 2 |
| Table 14.2-6.3 Raw cumulative incidence of MMR during re-treatment phase – Subset of Full Analysis Set entering the re-treatment phase |
| Table 14.2-6.4 Raw cumulative incidence of MMR during re-treatment phase , SDV sensitivity – Subset of Full Analysis Set entering the re-treatment phase222 |
| Table 14.2-7.1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase – Full Analysis Set |
| Table 14.2-7.1.1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase – LSC sub-study Full Analysis Set |
| Table 14.2-7.2 Raw cumulative incidence of MR 4.0 during post-randomization consolidation phase (ARM 2) – Subset of Full Analysis Set randomized to ARM 2 |
| Table 14.2-7.2.1 Raw cumulative incidence of MR 4.0 during post-randomization consolidation phase (ARM 2) – Subset of LSC sub-study Full Analysis Set randomized to ARM 2 |
| Table 14.2-7.3 Raw cumulative incidence of MR 4.0 during re-treatment phase – Subset of Full Analysis Set entering the re-treatment phase |
| Table 14.2-7.4 Raw cumulative incidence of MR 4.0 during re-treatment phase, SDV sensitivity – Subset of Full Analysis Set entering the re-treatment phase223 |
| Table 14.2-8.1 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase – Full Analysis Set |
| Table 14.2-8.1.1 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase – LSC sub-study Full Analysis Set |
| Table 14.2-8.2 Raw cumulative incidence of MR 4.5 during post-randomization consolidation phase (ARM 2) - Subset of Full Analysis Set randomized to Arm 2 |
| Table 14.2-8.2.1 Raw cumulative incidence of MR 4.5 during post-randomization consolidation phase (ARM 2) - Subset of LSC sub-study Full Analysis Set randomized to Arm 2 |
| Table 14.2-8.3 Raw cumulative incidence of MR 4.5 during re-treatment phase - Subset of Full Analysis Set entering the re-treatment phase |
| Table 14.2-8.4 Raw cumulative incidence of MR 4.5 during re-treatment phase, SDV sensitivity - Subset of Full Analysis Set entering the re-treatment phase225 |
| Table 14.2-9.1 Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase by halving time of BCR-ABL (IS) ratio – Full Analysis Set |

| Table 14.2-9.1.1 Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase by halving time of BCR-ABL (IS) ratio – LSC sub-study Full Analysis Set | 226 |
|---|---|
| Table 14.2-9.2 Raw cumulative incidence of MMR during post-randomization consolidation phase (ARM 2) by halving time of BCR-ABL (IS) ratio - Subset of Full Analysis Set randomized to Arm 2 | 227 |
| Table 14.2-9.2.1 Raw cumulative incidence of MMR during post-randomization consolidation phase (ARM 2) by halving time of BCR-ABL (IS) ratio - Subset of LSC sub-study Full Analysis Set randomized to Arm 2 | 228 |
| Table 14.2-9.3 Raw cumulative incidence of MMR during re-treatment phase by halving time of BCR-ABL (IS) ratio – Subset of Full Analysis Set entering the re-treatment phase | 228 |
| Table 14.2-10.1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase by halving time of BCR-ABL (IS) ratio – Full Analysis Set | 229 |
| Table 14.210.1.1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase by halving time of BCR-ABL (IS) ratio – LSC sub-study Full Analysis Set | 229 |
| Table 14.2-10.2 Raw cumulative incidence of MR 4.0 during post-randomization consolidation phase (ARM 2) by halving time of BCR-ABL (IS) ratio - Subset of Full Analysis Set randomized to Arm 2 | 229 |
| Table 14.2-10.2.1 Raw cumulative incidence of MR 4.0 during post-randomization consolidation phase (ARM 2) by halving time of BCR-ABL (IS) ratio - Subset of LSC sub-study Full Analysis Set randomized to Arm 2 | 229 |
| Table 14.2-10.3 Raw cumulative incidence of MR4.0 during re-treatment phase by halving time of BCR-ABL (IS) ratio – Subset of Full Analysis Set entering the re-treatment phase | 229 |
| Table 14.2-11.1 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase by halving time of BCR-ABL (IS) ratio – Full Analysis Set | 230 |
| Table 14.211.1.1 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase by halving time of BCR-ABL (IS) ratio – LSC sub-study Full Analysis Set | 230 |
| Table 14.2-11.2 Raw cumulative incidence of MR 4.5 during post-randomization consolidation phase (ARM 2) by halving time of BCR-ABL (IS) ratio - Subset of Full Analysis Set randomized to Arm 2 | 230 |
| Table14.2-11.2.1 Raw cumulative incidence of MR 4.5 during post-randomization consolidation phase (ARM 2) by halving time of BCR-ABL (IS) ratio - Subset of LSC sub-study Full Analysis Set randomized to Arm 2 | |
| Table 14.2-11.3 Raw cumulative incidence of MR4.5 during re-treatment phase by halving time of BCR-ABL (IS) ratio – Subset of Full Analysis Set entering the re-treatment phase | |
| Table 14.2-12.1 Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase by BCR-ABL (IS) ratio at Month 3 – Full | 231 |

| Table 14.2-12.1.1 Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase by BCR-ABL (IS) ratio at Month 3 – LSC sub-study Full Analysis Set | .231 |
|---|---|
| Table 14.2-12.2 Raw cumulative incidence of MMR during post-randomization consolidation phase (ARM 2) by BCR-ABL (IS) ratio at Month 3 - Subset of Full Analysis Set randomized to Arm 2 | .231 |
| Table 14.2-12.2.1 Raw cumulative incidence of MMR during post-randomization consolidation phase (ARM 2) by BCR-ABL (IS) ratio at Month 3 - Subset of LSC sub-study Full Analysis Set randomized to Arm 2 | .232 |
| Table 14.2-12.3 Raw cumulative incidence of MMR during re-treatment phase by BCR-ABL (IS) ratio at Month 3 – Subset of Full Analysis Set entering the retreatment phase | .232 |
| Table 14.2-13.1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase by BCR-ABL (IS) ratio at Month 3 – Full Analysis Set | .233 |
| Table 14.2-13.1.1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase by BCR-ABL (IS) ratio at Month 3 – LSC sub-study Full Analysis Set | .233 |
| Table 14.2-13.2 Raw cumulative incidence of MR 4.0 during post-randomization consolidation phase (ARM 2) by BCR-ABL (IS) ratio at Month 3 - Subset of Full Analysis Set randomized to Arm 2 | .233 |
| Table 14.2-13.2.1 Raw cumulative incidence of MR 4.0 during post-randomization consolidation phase (ARM 2) by BCR-ABL (IS) ratio at Month 3 - Subset of LSC sub-study Full Analysis Set randomized to Arm 2 | .233 |
| Table 14.2-13.3 Raw cumulative incidence of MR 4.0 during re-treatment phase by BCR-ABL (IS) ratio at Month 3 – Subset of Full Analysis Set entering the retreatment phase | .233 |
| Table 14.2-14.1 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase by BCR-ABL (IS) ratio at Month 3 – Full Analysis Set | .234 |
| Table 14.2-14.1.1 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase by BCR-ABL (IS) ratio at Month 3 – LSC sub-study Full Analysis Set | .234 |
| Table 14.2-14.2 Raw cumulative incidence of MR 4.5 during post-randomization consolidation phase (ARM 2) by BCR-ABL (IS) ratio at Month 3 - Subset of Full Analysis Set randomized to Arm 2 | .234 |
| Table 14.2-14.2.1 Raw cumulative incidence of MR 4.5 during post-randomization consolidation phase (ARM 2) by BCR-ABL (IS) ratio at Month 3 - Subset of LSC sub-study Full Analysis Set randomized to Arm 2 | .234 |
| Table 14.2-14.3 Raw cumulative incidence of MR 4.5 during re-treatment phase by BCR-ABL (IS) ratio at Month 3 – Subset of Full Analysis Set entering the retreatment phase | |
| Table 14.2-15.1 Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase by Sokal Risk category– Full Analysis Set | |
| Table 14.2-15.2 Raw cumulative incidence of MR4.0 during pre-randomization Induction/Consolidation phase by Sokal Risk category– Full Analysis Set | .235 |

| Table 14.2-15.3 Raw cumulative incidence of MR4.5 during pre-randomization Induction/Consolidation phase by Sokal Risk category—Full Analysis Set | .236 |
|---|---|
| Table 14.2-16.1 Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase by time since initial diagnosis of CML–Full Analysis Set | .237 |
| Table 14.2-16.2 Raw cumulative incidence of MR4.0 during pre-randomization Induction/Consolidation phase by time since initial diagnosis of CML – Full Analysis Set | .238 |
| Table 14.2-16.3 Raw cumulative incidence of MR4.5 during pre-randomization Induction/Consolidation phase by time since initial diagnosis of CML – Full Analysis Set | .238 |
| Table 14.2-17.1 Suboptimal response up to 24 months of pre-randomization Induction/Consolidation phase - Full Analysis Set patients who prematurely discontinued the pre-randomization Induction/Consolidation phase | .239 |
| Table 14.2-17.2 Suboptimal response up to 12 months of post-randomization Consolidation phase (ARM 2) - Subset of Full Analysis Set patients who prematurely discontinued the Induction/Consolidation phase randomized to Arm 2 | .240 |
| Table 14.2-18.1 Suboptimal response up to 24 months of pre-randomization Induction/Consolidation phase - Full Analysis Set | .240 |
| Table 14.2-18.2 Suboptimal response up to 12 months of post-randomization Consolidation phase - Subset of Full Analysis Set, randomized to ARM 2 | .240 |
| Table 14.2-19.1 Kinetics of BCR-ABL (IS) ratio during pre-randomization<br>Induction/Consolidation phase – Full Analysis Set | .241 |
| Table 14.2-19.1.1 Kinetics of BCR-ABL (IS) ratio during pre-randomization Induction/Consolidation phase – LSC sub-study Full Analysis Set | .241 |
| Table 14.2-19.2 Kinetics of BCR-ABL (IS) ratio during post-randomization consolidation phase (ARM 2) –Subset of Full Analysis Set randomized to Arm 2 | .242 |
| Table 14.2-19.2.1 Kinetics of BCR-ABL (IS) ratio during post-randomization consolidation phase (ARM 2) –Subset of LSC sub-study Full Analysis Set randomized to Arm 2 | .242 |
| Table 14.2-19.3 Kinetics of BCR-ABL (IS) ratio during TFR phase – Subset of Full Analysis Set entering the TFR phase | .243 |
| Table 14.2-19.4 Kinetics of BCR-ABL (IS) ratio during re-treatment phase – Subset of Full Analysis Set entering the re-treatment phase | .245 |
| Table 14.2-19.5 Kinetics of BCR-ABL (IS) ratio during TFR phase, SDV sensitivity – Subset of Full Analysis Set entering the TFR phase | .246 |
| Table 14.2-19.6 Kinetics of BCR-ABL (IS) ratio during re-treatment phase , SDV sensitivity – Subset of Full Analysis Set entering the re-treatment phase | .246 |
| Table 14.2-20.1 Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase - Full Analysis Set patients not reaching MMR at baseline | 247 |

| Table 14.2-20.2 Raw cumulative incidence of MMR during post-randomization Consolidation phase (ARM 2) - Subset of Full Analysis Set patients not reaching MMR at baseline, randomized to ARM 2 | .247 |
|---|---|
| Table 14.2-21.1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase - Full Analysis Set patients not reaching MR 4.0 at baseline | .247 |
| Table 14.2-21.2 Raw cumulative incidence of MR 4.0 during post-randomization Consolidation phase (ARM 2) - Subset of Full Analysis Set patients not reaching MR 4.0 at baseline, randomized to ARM 2 | .247 |
| Table 14.2-22.1 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase - Full Analysis Set patients not reaching MR 4.5 at baseline | .247 |
| Table 14.2-22.2 Raw cumulative incidence of MR 4.5 during post-randomization Consolidation phase (ARM 2) - Subset of Full Analysis Set patients not reaching MR 4.5 at baseline, randomized to ARM 2 | .248 |
| Table 14.2-22.3 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase - Full Analysis Set patients not reaching MMR at baseline | .248 |
| Table 14.2-22.4 Raw cumulative incidence of MR 4.0 during post-randomization Consolidation phase (ARM 2) - Subset of Full Analysis Set patients not reaching MMR at baseline, randomized to ARM 2 | .248 |
| Table 14.2-22.5 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase - Full Analysis Set patients not reaching MMR at baseline | .248 |
| Table 14.2-22.6 Raw cumulative incidence of MR 4.5 during post-randomization Consolidation phase (ARM 2) - Subset of Full Analysis Set patients not reaching MMR at baseline, randomized to ARM 2 | .248 |
| Table 14.2-23.1 Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase by BCR-ABL(IS) ratio at baseline - Full Analysis Set | .249 |
| Table 14.2-23.1.1 Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase by BCR-ABL (IS) ratio at baseline– LSC substudy Full Analysis Set | .250 |
| Table 14.2-23.2 Raw cumulative incidence of MMR during post-randomization consolidation phase (ARM 2) by BCR-BL(IS) ratio at baseline - Subset of Full Analysis Set, randomized to ARM 2 | .250 |
| Table 14.2-23.2.1 Raw cumulative incidence of MMR during post-randomization consolidation phase (ARM 2) by BCR-BL(IS) ratio at baseline - Subset of LSC sub-study Full Analysis Set, randomized to ARM 2 | |
| Table 14.2-23.3 Raw cumulative incidence of MMR during re-treatment phase by BCR-BL(IS) ratio at baseline – Subset of Full Analysis Set entering the retreatment phase | |
| Table 14.2-24.1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase by BCR-ABL(IS) ratio at baseline - Full Analysis Set | .252 |

| Table 14.2-24.1.1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase by BCR-ABL (IS) ratio at baseline– LSC substudy Full Analysis Set | 252 |
|---|---|
| Table 14.2-24.2 Raw cumulative incidence of MR 4.0 during post-randomization consolidation phase (ARM 2) by BCR-BL(IS) ratio at baseline - Subset of Full Analysis Set, randomized to ARM 2 | 252 |
| Table 14.2-24.2.1 Raw cumulative incidence of MR 4.0 during post-randomization consolidation phase (ARM 2) by BCR-BL(IS) ratio at baseline - Subset of LSC sub-study Full Analysis Set , randomized to ARM 2 | 252 |
| Table 14.2-24.3 Raw cumulative incidence of MR 4.0 during re-treatment phase by BCR-BL(IS) ratio at baseline – Subset of Full Analysis Set entering the retreatment phase | 252 |
| Table 14.2-25.1 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase by BCR-ABL(IS) ratio at baseline - Full Analysis Set | 253 |
| Table 14.2-25.1.1 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase by BCR-ABL (IS) ratio at baseline– LSC substudy Full Analysis Set | 253 |
| Table 14.2-25.2 Raw cumulative incidence of MR 4.5 during post-randomization consolidation phase (ARM 2) by BCR-BL(IS) ratio at baseline - Subset of Full Analysis Set, randomized to ARM 2 | 253 |
| Table 14.2-25.2.1 Raw cumulative incidence of MR 4.5 during post-randomization consolidation phase (ARM 2) by BCR-BL(IS) ratio at baseline - Subset of LSC sub-study Full Analysis Set, randomized to ARM 2 | 253 |
| Table 14.2-25.3 Raw cumulative incidence of MR 4.5 during re-treatment phase by BCR-BL(IS) ratio at baseline – Subset of Full Analysis Set entering the retreatment phase | 253 |
| Table 14.2-26.1 Raw cumulative loss of MMR during TFR phase –Subset of Full | 254 |
| Table 14.2-26.2 Raw cumulative loss of MR4.0 during TFR phase –Subset of Full Analysis Set entering the TFR phase | 255 |
| Table 14.2-26.3 Raw cumulative loss of MR4.5 during TFR phase –Subset of Full Analysis Set entering the TFR phase with MR4.5 | 255 |
| Table 14.2-26.4 Raw cumulative loss of MMR during TFR phase, SDV sensitivity – Subset of Full Analysis Set entering the TFR phase | 256 |
| Table 14.2-26.5 Raw cumulative loss of MR4.0 during TFR phase, SDV sensitivity —Subset of Full Analysis Set entering the TFR phase | 256 |
| Table 14.2-26.6 Raw cumulative loss of MR4.5 during TFR phase, SDV sensitivity -Subset of Full Analysis Set entering the TFR phase with MR4.5 | 256 |
| Table 14.2-27.1 Descriptive Statistics for CD34 cells: Total percentage – LSC substudy Full Analysis Set | 257 |
| Table 14.2-28.1 Descriptive Statistics for CD34+/CD38+ cells: Percentage from total CD34+ cells – LSC sub-study Full Analysis Set | 259 |
| Table 14.2-28.2 Descriptive Statistics for number of events sorted in CD34+/CD38+ cells – LSC sub-study Full Analysis Set | 260 |

| Table 14.2-28.3 Ph+ by HIS status, in CD34+/CD38+ cells – LSC sub-study Full Analysis Set |
|---|
| Table 14.2-28.4 Descriptive statistics of Ph+ in CD34+/CD38+ cells- LSC sub-study Full Analysis Set |
| Table 14.2-28.5 BCR-ABL by RT-PCR status, in CD34+/CD38+ cells – LSC substudy Full Analysis Set |
| Table 14.2-29.1 Descriptive Statistics for CD34+/CD38- cells: Percentage from total CD34+ cells – LSC sub-study Full Analysis Set |
| Table 14.2-29.2 Descriptive Statistics for number of events sorted in CD34+/CD38-cells – LSC sub-study Full Analysis Set |
| Table 14.2-29.3 Ph+ by HIS status, in CD34+/CD38- cells – LSC sub-study Full Analysis Set |
| Table 14.2-29.4 Descriptive statistics of Ph+ in CD34+/CD38- cells– LSC sub-study Full Analysis Set |
| Table 14.2-29.5 BCR-ABL by RT-PCR status, in CD34+/CD38- cells – LSC substudy Full Analysis Set |
| Table 14.2-30.1 Descriptive Statistics for Immunophenotypically aberrant CD34+ cells: Percentage from total CD34+ cells –LSC sub-study Full Analysis Set263 |
| Table 14.2-30.2 Descriptive Statistics for number of events sorted in Immunophenotypically aberrant CD34+ cells – LSC sub-study Full Analysis Set |
| Table 14.2-30.3 Ph+ by HIS status, in Immunophenotypically aberrant CD34+ cells - LSC sub-study Full Analysis Set |
| Table 14.2-30.4 Descriptive statistics of Ph+ in Immunophenotypically aberrant CD34+ cells– LSC sub-study Full Analysis Set |
| Table 14.2-30.5 BCR-ABL by RT-PCR status, in Immunophenotypically aberrant CD34+ cells – LSC sub-study Full Analysis Set |
| Table 14.2-31.1 Descriptive Statistics for Immunophenotypically aberrant CD34-cells: Percentage from total CD34+ cells – LSC sub-study Full Analysis Set264 |
| Table 14.2-31.2 Descriptive Statistics for number of events sorted in Immunophenotypically aberrant CD34- cells- LSC sub-study Full Analysis Set |
| Table 14.2-31.3 Ph+ by HIS status, in Immunophenotypically aberrant CD34- cells – LSC sub-study Full Analysis Set |
| Table 14.2-31.4 Descriptive statistics of Ph+ in Immunophenotypically aberrant CD34- cells– LSC sub-study Full Analysis Set |
| Table 14.2-31.5 BCR-ABL by RT-PCR status, in Immunophenotypically aberrant CD34- cells – LSC sub-study Full Analysis Set |
| Table 14.2-32.1 Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase by duration of prior exposure to Imatinib - Full Analysis Set |
| Table 14.2-32.1.1 Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase by by prior Imatib treatment duration – LSC sub-study Full Analysis Set |

| Table 14.2-32.2 Raw cumulative incidence of MMR during post-randomization consolidation phase (ARM 2) by prior Imatib treatment duration - Subset of Full Analysis Set, randomized to ARM 2 | 266 |
|---|---|
| Table 14.2-32.2.1 Raw cumulative incidence of MMR during post-randomization consolidation phase (ARM 2) by prior Imatib treatment duration - Subset of LSC sub-study Full Analysis Set , randomized to ARM 2 | 267 |
| Table 14.2-32.3 Raw cumulative incidence of MMR during re-treatment phase by prior Imatib treatment duration – Subset of Full Analysis Set entering the retreatment phase | 267 |
| Table 14.2-33.1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase by prior Imatib treatment duration - Full Analysis Set | 268 |
| Table 14.2-33.1.1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase by prior Imatib treatment duration – LSC substudy Full Analysis Set | 268 |
| Table 14.2-33.2 Raw cumulative incidence of MR 4.0 during post-randomization consolidation phase (ARM 2) by prior Imatib treatment duration - Subset of Full Analysis Set, randomized to ARM 2 | 268 |
| Table 14.2-33.2.1 Raw cumulative incidence of MR 4.0 during post-randomization consolidation phase (ARM 2) by prior Imatib treatment duration - Subset of LSC sub-study Full Analysis Set , randomized to ARM 2 | 268 |
| Table 14.2-33.3 Raw cumulative incidence of MR 4.0 during re-treatment phase by prior Imatib treatment duration – Subset of Full Analysis Set entering the retreatment phase | 268 |
| Table 14.2-34.1 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase by prior Imatib treatment duration - Full Analysis Set | 269 |
| Table 14.2-34.1.1 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase by prior Imatib treatment duration – LSC sub- | 269 |
| Table 14.2-34.2 Raw cumulative incidence of MR 4.5 during post-randomization consolidation phase (ARM 2) by prior Imatib treatment duration - Subset of Full Analysis Set, randomized to ARM 2 | 269 |
| Table 14.2-34.2.1 Raw cumulative incidence of MR 4.5 during post-randomization consolidation phase (ARM 2) by prior Imatib treatment duration - Subset of LSC sub-study Full Analysis Set , randomized to ARM 2 | 269 |
| Table 14.2-34.3 Raw cumulative incidence of MR 4.5 during re-treatment phase by prior Imatib treatment duration – Subset of Full Analysis Set entering the retreatment phase | 269 |
| Section 14.3 – Safety data | |
| Table 14.3-1.1 Duration of exposure to study treatment during pre-randomization | 271 |
| Table 14.3-1.1.1 Duration of exposure to study treatment during pre-randomization Induction/Consolidation— LSC sub-study Safety Set | |

| Table 14.3-1.2 Duration of exposure to study treatment during post-randomization Consolidation phase (ARM 2) - Subset of Safety Set randomized to Arm 2 | 272 |
|---|---|
| Table 14.3-1.2.1 Duration of exposure to study treatment during post-randomization Consolidation phase (ARM 2) - Subset of LSC sub-study Safety Set randomized to Arm 2 | .272 |
| Table 14.3-1.1.3 Duration of exposure to study treatment during re-treatment phase – Subset of Safety Set entering the re-treatment phase | |
| Table 14.3-1.1.21 Duration of exposure to study treatment during pre-randomization Induction/Consolidation phase, by stable MR4.0 at 24 months and halving time - Safety Set | 273 |
| Table 14.3-1.1.22 Duration of exposure to study treatment during pre-randomization Induction/Consolidation phase, by stable MR4.0 by 24 months and halving time - Safety Set | 275 |
| Table 14.3-2.1 Relative dose intensity and average daily dose during pre-<br>randomization Induction/Consolidation phase – Safety Set | 276 |
| Table 14.3-2.1.1 Relative dose intensity and average daily dose during pre-<br>randomization Induction/Consolidation phase – LSC sub-study Safety Set | .277 |
| Table 14.3-2.2 Relative dose intensity and average daily dose during post-randomization consolidation phase (ARM 2) – Subset of Safety Set randomized to Arm 2 | .277 |
| Table 14.3-2.2.1 Relative dose intensity and average daily dose during post-<br>randomization consolidation phase (ARM 2) – Subset of LSC sub-study<br>Safety Set randomized to Arm 2 | 277 |
| Table 14.3-2.3 Relative dose intensity and average daily dose during re-treatment phase – Subset of Safety Set entering the re-treatment phase | .278 |
| Table 14.3-3.1 Dose reduction and interruption during pre-randomization Induction/Consolidation phase - Safety Set | .279 |
| Table 14.3-3.1.1 Dose reduction and interruption during pre-randomization Induction/Consolidation phase – LSC sub-study Safety Set | 279 |
| Table 14.3-3.2 Dose reduction and interruption during post-randomization consolidation phase (ARM 2) – Subset of Safety Set randomized to Arm 2 | .280 |
| Table 14.3-3.2.1 Dose reduction and interruption during post-randomization consolidation phase (ARM 2) – Subset of LSC sub-study Safety Set randomized to Arm 2 | .280 |
| Table 14.3-3.3 Dose reduction and interruption during re-treatment phase – Subset of Safety Set entering the re-treatment phase | |
| Table 14.3-4.1 Concomitant medication by ATC class and preferred term during prerandomization Induction/Consolidation phase Full Analysis Set | |
| Table 14.3-4.1.1 Concomitant medication by ATC class and preferred term during pre-randomization Induction/Consolidation phase LSC sub-study Full Analysis Set | 282 |
| Table 14.3-4.2 Concomitant medication by ATC class and preferred term during post-randomization consolidation phase (ARM 2)— Subset of Full Analysis Set randomized to Arm 2 | 283 |

| Table 14.3-4.2.1 Concomitant medication by ATC class and preferred term during post-randomization consolidation phase (ARM 2)— Subset of LSC sub-study Full Analysis Set randomized to Arm 2 | .284 |
|---|---|
| Table 14.3-4.3 Concomitant medication by ATC class and preferred term during TFR phase – Subset of Full Analysis Set entering the TFR phase | .285 |
| Table 14.3-4.4 Concomitant medication by ATC class and preferred term during retreatment phase – Subset of Full Analysis Set entering the re-treatment phase | 286 |
| Table 14.3-5.1.1 Hematology shift table based on CTCAE grade during Pre-<br>Randomization pre-randomization Induction/Consolidation –Full Analysis<br>Set | .287 |
| Table 14.3-5.1.2 Hematology shift table based on CTCAE grade during post-randomization consolidation phase (ARM 2)— Subset of Full Analysis Set randomized to Arm 2 | .289 |
| Table 14.3-5.1.3 Hematology shift table based on CTCAE grade during re-treatment phase – Subset of Full Analysis Set entering the re-treatment phase | .290 |
| Table 14.3-5.1.4 Hematology shift table based on CTCAE grade during whole study period – Full Analysis Set | .292 |
| Table 14.3-5.1.5 Hematology shift table based on CTCAE grade during re-treatment phase, SDV sensitivity — Subset of Full Analysis Set entering the retreatment phase | .293 |
| Table 14.3-5.1.6 Hematology shift table based on CTCAE grade during whole study period, SDV sensitivity– Full Analysis Set | .293 |
| Table 14.3-5.2.1 Biochemistry shift table based on CTCAE grade during post-randomization consolidation phase (ARM 2)— Subset of Full Analysis Set randomized to Arm 2 | .294 |
| Table 14.3-5.2.2 Biochemistry shift table based on CTCAE grade during retreatment phase—Subset of Full Analysis Set entering the re-treatment phase | .294 |
| Table 14.3-5.2.3 Biochemistry shift table based on CTCAE grade during whole study period – Full Analysis Set | .294 |
| Table 14.3-5.2.4 Biochemistry shift table based on CTCAE grade during retreatment phase, SDV sensitivity— Subset of Full Analysis Set entering the retreatment phase | .294 |
| Table 14.3-5.2.5 Biochemistry shift table based on CTCAE grade during whole study period, SDV sensitivity – Full Analysis Set | .294 |
| Table 14.3-6.1.1 Hematology shift table based on normal range for parameters with no defined CTCAE grades during post-randomization consolidation phase (ARM 2)— Subset of Full Analysis Set randomized to Arm 2 | .295 |
| Table 14.3-6.1.2 Hematology shift table based on normal range for parameters with no defined CTCAE grades during re-treatment phase – Subset of Full Analysis Set entering the re-treatment phase | .296 |
| Table 14.3-6.1.3 Hematology shift table based on normal range for parameters with no defined CTCAE grades during whole study period –Full Analysis Set | .297 |
| Table 14.3-6.1.4 Hematology shift table based on normal range for parameters with no defined CTCAE grades during re-treatment phase, SDV sensitivity – Subset of Full Analysis Set entering the re-treatment phase | .298 |
| , r | _ |
| Table 14.3-6.1.5 Hematology shift table based on normal range for parameters with no defined CTCAE grades during whole study period, SDV sensitivity –Full Analysis Set | 298 |
|---|---|
| Table 14.3-6.2.1 Biochemistry shift table based on normal range for parameters with no defined CTCAE grades during post-randomization consolidation phase (ARM 2) – Subset of Full Analysis Set randomized to Arm 2 | .299 |
| Table 14.3-6.2.2 Biochemistry shift table based on normal range for parameters with no defined CTCAE grades during re-treatment phase – Subset of Full Analysis Set entering the re-treatment phase | .299 |
| Table 14.3-6.2.3 Biochemistry shift table based on normal range for parameters with no defined CTCAE grades during whole study period –Full Analysis Set | 299 |
| Table 14.3-6.2.4 Biochemistry shift table based on normal range for parameters with no defined CTCAE grades during re-treatment phase, SDV sensitivity – Subset of Full Analysis Set entering the re-treatment phase | .299 |
| Table 14.3-6.2.5 Biochemistry shift table based on normal range for parameters with no defined CTCAE grades during whole study period, SDV sensitivity –Full Analysis Set | .299 |
| Table 14.3-7.1 ECG shift table based on notable values during Pre-randomization Induction Consolidation–Full Analysis Set | .300 |
| Table 14.3-7.2 ECG shift table based on notable values during post-randomization consolidation phase (ARM 2) – Subset of Full Analysis Set randomized to Arm 2 | .301 |
| Table 14.3-7.3 ECG shift table based on notable values during re-treatment phase – Subset of Full Analysis Set entering the re-treatment phase | 302 |
| Table 14.3-7.4 Notable ECG values during pre-randomization Ind/Cons –Full Analysis Set | .303 |
| Table 14.3-7.5 Notable ECG values during post-randomization consolidation phase (ARM 2)— Subset of Full Analysis Set randomized to Arm 2 | .304 |
| Table 14.3-7.6 Notable ECG values during re-treatment phase – Subset of Full Analysis Set entering the re-treatment phase | .305 |
| Table 14.3-7.7 ECG shift table based on notable values during re-treatment phase, SDV sensitivity – Subset of Full Analysis Set entering the re-treatment phase. | .305 |
| Table 14.3-7.8 Notable ECG values during re-treatment phase, SDV sensitivity – Subset of Full Analysis Set entering the re-treatment phase | .305 |
| Table 14.3-8.1 Echocardiography assessment at baseline – Full Analysis Set | .306 |
| Table 14.3-8.2 Echocardiography shift table based on overall interpretation - Full Analysis Set | .307 |
| Table 14.3-8.3 Echocardiography shift table based on overall interpretation, SDV sensitivity - Full Analysis Set | .308 |
| Table 14.3-9.1 Summary statistics of total cholesterol, HDL, LDL, glucose, microalbumin and HbA1c over Induction/Consolidation phase – Full Analysis Set | 309 |
| Table 14.3-9.2.1 Total cholesterol shift table based on specific levels during Induction Consolidation – Full Analysis Set | 310 |

| Table 14.3-9.2.2 Total cholesterol shift table based on specific levels during TFR phase – Subset of Full Analysis Set entering the TFR phase | 311 |
|---|---|
| Table 14.3-9.2.3 Total cholesterol shift table based on specific levels during Retreatment phase — Subset of Full Analysis Set entering the Re-treatment phase | 311 |
| Table 14.3-9.2.4 Total cholesterol shift table based on specific levels during TFR phase, SDV sensitivity – Subset of Full Analysis Set entering the TFR phase | 311 |
| Table 14.3-9.2.5 Total cholesterol shift table based on specific levels during Retreatment phase, SDV sensitivity – Subset of Full Analysis Set entering the Re-treatment phase | 312 |
| Table 14.3-10.1.1 Fasting glucose shift table based on specific levels during Induction Consolidation – Full Analysis Set | 313 |
| Table 14.3-10.1.2 Fasting glucose shift table based on specific levels during TFR phase — Subset of Full Analysis Set entering the TFR phase | 314 |
| Table 14.3-10.1.3 Fasting glucose shift table based on specific levels during Retreatment phase — Subset of Full Analysis Set entering the Re-treatment phase | 314 |
| Table 14.3-10.1.4 Fasting glucose shift table based on specific levels during TFR phase, SDV sensitivity – Subset of Full Analysis Set entering the TFR phase. | 314 |
| Table 14.3-10.1.5 Fasting glucose shift table based on specific levels during Retreatment phase, SDV sensitivity — Subset of Full Analysis Set entering the Re-treatment phase | 315 |
| Table 14.3-11.1 Vital Signs during Induction Consolidation – Full Analysis Set | 316 |
| Table 14.3-11.2 Vital Signs during TFR phase – Subset of Full Analysis Set entering the TFR phase | 319 |
| Table 14.3-11.3 Vital Signs during Re-treatment phase — Subset of Full Analysis Set entering the Re-treatment phase | 319 |
| Table 14.3-11.4 Vital Signs during TFR phase, SDV sensitivity – Subset of Full Analysis Set entering the TFR phase | 320 |
| Table 14.3-11.5 Vital Signs during Re-treatment phase, SDV sensitivity – Subset of Full Analysis Set entering the Re-treatment phase | 320 |
| Table 14.3-12.1 Survival follow-up – Full Analysis Set | 321 |
| Table 14.3-12.2 Survival follow-up, SDV sensitivity – Full Analysis Set | 322 |
| Table 14.3-13.1 Safety follow-up – Full analysis Set | 323 |
| Table 14.3-13.2 Safety follow-up, SDV sensitivity – Full analysis Set | 323 |
| Section 14.3.1 – Displays of adverse events | 324 |
| Figure 14.3.1-1.1 Kaplan-Meier analysis of time-to-first CVEs during the pre-<br>randomization Induction/Consolidation phase – Full Analysis Set | 324 |
| Figure 14.3.1-1.2 Kaplan-Meier analysis of time-to-first CVEs during the post-randomization consolidation phase (ARM 2) – Subset of Full Analysis Set randomized to Arm 2 | 325 |
| Figure 14.3.1-1.3 Kaplan-Meier analysis of time-to-first CVEs during the the TFR phase – Subset of Full Analysis Set entering the TFR phase | 326 |

| Figure | 14.3.1-1.4 Kaplan-Meier analysis of time-to-first CVEs during the retreatment phase – Subset of Full Analysis Set entering the re-treatment phase | 326 |
|---|---|---|
| Figure | 14.3.1-2.1 Number of sorted events by HIS CD34+/CD38+ cells | 327 |
| Figure | 14.3.1-2.2 Number of sorted events by PCR CD34+/CD38+ cells | 328 |
| Figure | 14.3.1-3.1 Number of sorted events by HIS CD34+/CD38- cells | 328 |
| Figure | 14.3.1-3.2 Number of sorted events by PCR CD34+/CD38- cells | 328 |
| Figure | 14.3.1-4.1 Number of sorted events by HIS Immunophenotypically aberrant CD34+ cells | .328 |
| Figure | 14.3.1-4.2 Number of sorted events by PCR Immunophenotypically aberrant CD34+ cells | .328 |
| Figure | 14.3.1-5.1 Number of sorted events by HIS Immunophenotypically aberrant CD34- cells | .328 |
| Figure | 14.3.1-5.2 Number of sorted events by PCR Immunophenotypically aberrant CD34- cells | .328 |
| Figure | 14.3.1-6.1 Number of HIS+ subjects CD34+/CD38+ cells – LSC substudy Full Analysis Set | .329 |
| Figure | 14.3.1-6.2 Number of PCR subjects CD34+/CD38+ cells – LSC substudy Full Analysis Set | .330 |
| _ | 14.3.1-7.1 Number of HIS+ subjects CD34+/CD38- cells – LSC substudy Full Analysis Set | .330 |
| Figure | 14.3.1-7.2 Number of PCR subjects CD34+/CD38- cells – LSC substudy Full Analysis Set | .330 |
| Figure | 14.3.1-8.1 Number of HIS+ subjects Immunophenotypically aberrant CD34+ cells – LSC substudy Full Analysis Set | .330 |
| Figure | 14.3.1-8.2 Number of PCR subjects Immunophenotypically aberrant CD34+ cells – LSC substudy Full Analysis Set | .330 |
| Figure | 14.3.1-9.1 Number of HIS+ subjects Immunophenotypically aberrant CD34-cells – LSC substudy Full Analysis Set | .330 |
| Figure | 14.3.1-9.2 Number of PCR subjects Immunophenotypically aberrant CD34-cells – LSC substudy FAS | .330 |
| Figure | 14.3.1-10 Number of patients with detectable LSC – LSC substudy Full Analysis Set | .331 |
| Table 1 | 14.3.1-1.1 Overall summary of treatment-emergent adverse events occurring during pre-randomization Induction/consolidation phase – Full Analysis Set | .332 |
| Table 1 | 14.3.1-1.2 Overall summary of treatment-emergent adverse events occurring during post-randomization consolidation phase (ARM 2) – Subset of Full Analysis Set randomized to Arm 2 | .334 |
| Table 1 | 14.3.1-1.3 Overall summary of treatment-emergent adverse events occurring during re-treatment phase — Subset of Full Analysis Set entering the retreatment phase | .336 |
| Table 1 | 14.3.1-1.4 Overall summary of adverse events occurring during TFR phase – Subset of Full Analysis Set entering the TFR phase | .337 |

| Table 14.3.1-2.1 Overall summary of frequent [1] treatment-emergent adverse events occurring during pre-randomization Induction/consolidation phase – Full Analysis Set | .338 |
|---|---|
| Table 14.3.1-2.2 Overall summary of frequent [1] treatment-emergent adverse events occurring during post-randomization consolidation phase (ARM 2) – Subset of Full Analysis Set randomized to Arm 2 | |
| Table 14.3.1-2.3 Overall summary of frequent [1] treatment-emergent adverse events occurring during re-treatment phase — Subset of Full Analysis Set entering the re-treatment phase | .338 |
| Table 14.3.1-2.4 Overall summary of frequent [1] adverse events occurring during TFR phase – Subset of Full Analysis Set entering the TFR phase | .339 |
| Table 14.3.1-3.1.1 Treatment Emergent adverse events incidence, regardless of study drug relationship, occurring during pre-randomization Induction/consolidation phase by system organ class and preferred term - overall and maximum grade 3/4 – Full Analysis Set | .340 |
| Table 14.3.1-3.1.2 Treatment Emergent adverse events occurence, regardless of study drug relationship, occurring during pre-randomization Induction/consolidation phase by system organ class and preferred term - overall and maximum grade 3/4 – Full Analysis Set | .341 |
| Table 14.3.1-3.2.1 Treatment Emergent adverse events incidence, regardless of study drug relationship, occurring during post-randomization consolidation phase (ARM 2) by system organ class and preferred term - overall and maximum grade 3/4 – Subset of Full Analysis Set randomized to Arm 2 | .342 |
| Table 14.3.1-3.2.2 Treatment Emergent adverse events occurence, regardless of study drug relationship, occurring during post-randomization consolidation phase (ARM 2) by system organ class and preferred term - overall and maximum grade 3/4 – Subset of Full Analysis Set randomized to Arm 2 | .343 |
| Table 14.3.1-3.3.1 Treatment-emergent adverse events incidence, regardless of study drug relationship, by system organ class and preferred term during retreatment phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the re-treatment phase | .344 |
| Table 14.3.1-3.3.2 Treatment-emergent adverse events occurrence, regardless of study drug relationship, by system organ class and preferred term during retreatment phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the re-treatment phase | .345 |
| Table 14.3.1-3.4.1 Adverse events incidence, regardless of study drug relationship, by system organ class and preferred term during TFR phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the TFR phase | .345 |
| Table 14.3.1-3.4.2 Adverse events occurrence, regardless of study drug relationship, by system organ class and preferred term during TFR phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the TFR phase | .345 |
| Table 14.3.1-3.5.1 Frequent [1] Treatment Emergent adverse events incidence, regardless of study drug relationship occurring during pre-randomization Induction/consolidation phase by system organ class and preferred term | 246 |
| overall and maximum grade 3/4 – Full Analysis Set | .346 |

| Table 14.3.1-3.5.2 Frequent [1] Treatment Emergent adverse events incidence, regardless of study drug relationship occurring during post-randomization consolidation phase (ARM 2) by system organ class and preferred termoverall and maximum grade 3/4 – Subset of Full Analysis Set randomized to Arm 2 | 346 |
|---|---|
| Table 14.3.1-3.5.3 Frequent [1] Treatment Emergent adverse events incidence, regardless of study drug relationship occurring during re-treatment phase by system organ class and preferred term- overall and maximum grade 3/4 — Subset of Full Analysis Set entering the re-treatment phase | 347 |
| Table 14.3.1-3.5.4 Frequent [1] adverse events incidence, regardless of study drug relationship occurring during TFR phase by system organ class and preferred term - overall and maximum grade 3/4 – Subset of Full Analysis Set entering the TFR phase | |
| Table 14.3.1-4.1.1 Serious treatment-emergent adverse events incidence, regardless of study drug relationship, by system organ class and preferred term during pre-randomization Induction/consolidation phase – overall and maximum grade 3/4 –Full Analysis Set | 348 |
| Table 14.3.1-4.1.2 Serious treatment-emergent adverse events occurence, regardless of study drug relationship, by system organ class and preferred term during pre-randomization Induction/consolidation phase – overall and maximum grade 3/4 –Full Analysis Set | 348 |
| Table 14.3.1-4.2.1 Serious treatment-emergent adverse events incidence, regardless of study drug relationship, by system organ class and preferred term during post-randomization consolidation phase (ARM 2) – overall and maximum grade 3/4 – Subset of Full Analysis Set randomized to Arm 2 | 349 |
| Table 14.3.1-4.2.2 Serious treatment-emergent adverse events occurrence, regardless of study drug relationship, by system organ class and preferred term during post-randomization consolidation phase (ARM 2) – overall and maximum grade 3/4 – Subset of Full Analysis Set randomized to Arm 2 | 349 |
| Table 14.3.1-4.3.1 Serious treatment-emergent adverse events incidence, regardless of study drug relationship, by system organ class and preferred term during re-treatment phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the re-treatment phase | 350 |
| Table 14.3.1-4.3.2 Serious treatment-emergent adverse events occurrence, regardless of study drug relationship, by system organ class and preferred term during re-treatment phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the re-treatment phase | |
| Table 14.3.1-4.4.1 Serious adverse events incidence, regardless of study drug relationship, by system organ class and preferred term during TFR phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the TFR phase | 350 |
| Table 14.3.1-4.4.2 Serious adverse events occurence, regardless of study drug relationship, by system organ class and preferred term during TFR phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the TFR phase | |
| Table 14.3.1-4.5.1 Frequent [1] Serious Treatment Emergent adverse events incidence, regardless of study drug relationship occurring during pre- | |

| randomization Induction/consolidation phase by system organ class and preferred term - overall and maximum grade 3/4 – Full Analysis Set351 |
|---|
| Table 14.3.1-4.5.2 Frequent [1] Serious Treatment Emergent adverse events incidence, regardless of study drug relationship occurring during post-randomization consolidation phase (ARM 2) by system organ class and preferred term - overall and maximum grade 3/4 – Subset of Full Analysis Set randomized to Arm 2 |
| Table 14.3.1-4.5.3 Frequent [1] Serious Treatment Emergent adverse events incidence, regardless of study drug relationship occurring during re-treatment phase by system organ class and preferred term - overall and maximum grade 3/4 – Subset of Full Analysis Set entering the re-treatment phase |
| Table 14.3.1-4.5.4 Frequent [1] Serious adverse events incidence, regardless of study drug relationship occurring during TFR phase by system organ class and preferred term - overall and maximum grade 3/4 – Subset of Full Analysis Set entering the TFR phase |
| Table 14.3.1-4.6.1 Serious treatment-emergent adverse events incidence, suspected to be study drug related, by system organ class and preferred term during prerandomization Induction/consolidation phase – overall and maximum grade 3/4 –Full Analysis Set |
| Table 14.3.1-4.6.2 Serious treatment-emergent adverse events occurence, suspected to be study drug related, by system organ class and preferred term during prerandomization Induction/consolidation phase – overall and maximum grade 3/4 –Full Analysis Set |
| Table 14.3.1-4.7.1 Serious treatment-emergent adverse events incidence, suspected to be study drug related, by system organ class and preferred term during post-randomization consolidation phase (ARM 2) – overall and maximum grade 3/4 – Subset of Full Analysis Set randomized to Arm 2 |
| Table 14.3.1-4.7.2 Serious treatment-emergent adverse events occurrence, suspected to be study drug related, by system organ class and preferred term during post-randomization consolidation phase (ARM 2) – overall and maximum grade 3/4 – Subset of Full Analysis Set randomized to Arm 2 |
| Table 14.3.1-4.8.1 Serious treatment-emergent adverse events incidence, suspected to be study drug related, by system organ class and preferred term during retreatment phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the re-treatment phase |
| Table 14.3.1-4.8.2 Serious treatment-emergent adverse events occurrence, suspected to be study drug related, by system organ class and preferred term during retreatment phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the re-treatment phase |
| Table 14.3.1-4.9.1 Serious adverse events incidence, suspected to be study drug related, by system organ class and preferred term during TFR phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the TFR phase |
| Table 14.3.1-4.9.2 Serious adverse events occurrence, suspected to be study drug related, by system organ class and preferred term during TFR phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the TFR phase |

| Table 14.3.1-5.1.1 Treatment-emergent adverse events incidence leading to study drug discontinuation by system organ class and preferred term during prerandomization Induction/Consolidation phase – overall and maximum grade 3/4 –Full Analysis Set | .354 |
|---|---|
| Table 14.3.1-5.1.2 Treatment-emergent adverse events occurence leading to study drug discontinuation by system organ class and preferred term during prerandomization Induction/Consolidation phase – overall and maximum grade 3/4 –Full Analysis Set | .355 |
| Table 14.3.1-5.2.1 Treatment-emergent adverse events incidence leading to study drug discontinuation by system organ class and preferred term during post-randomization phase (ARM 2) – overall and maximum grade 3/4 – Subset of Full Analysis Set randomized to Arm 2 | .355 |
| Table 14.3.1-5.2.2 Treatment-emergent adverse events occurrence leading to study drug discontinuation by system organ class and preferred term during post-randomization phase (ARM 2)— overall and maximum grade 3/4 — Subset of Full Analysis Set randomized to Arm 2 | .355 |
| Table 14.3.1-5.3.1 Treatment-emergent adverse events incidence leading to study drug discontinuation by system organ class and preferred term during retreatment phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the re-treatment phase | .356 |
| Table 14.3.1-5.3.2 Treatment-emergent adverse events occurrence leading to study drug discontinuation by system organ class and preferred term during retreatment phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the re-treatment phase | .356 |
| Table 14.3.1-6.1.1 Treatment-emergent adverse events incidence requiring dosage adjustment or temporarily interruption by system organ class and preferred term during pre-randomization Induction/ consolidation phase — overall and maximum grade 3/4—Full Analysis Set | .356 |
| Table 14.3.1-6.1.2 Treatment-emergent adverse events occurrence requiring dosage adjustment or temporarily interruption by system organ class and preferred term during pre-randomization Induction/consolidation phase – overall and maximum grade 3/4 –Full Analysis Set | .357 |
| Table 14.3.1-6.2.1 Treatment-emergent adverse events incidence requiring dosage adjustment or temporarily interruption by system organ class and preferred term during post-randomization consolidation phase (ARM 2) – overall and maximum grade 3/4 – Subset of Full Analysis Set randomized to Arm 2 | .357 |
| Table 14.3.1-6.2.2 Treatment-emergent adverse events occurrence requiring dosage adjustment or temporarily interruption by system organ class and preferred term during post-randomization consolidation phase (ARM 2) – overall and maximum grade 3/4 – Subset of Full Analysis Set randomized to Arm 2 | .357 |
| Table 14.3.1-6.3.1 Treatment-emergent adverse events incidence requiring dosage adjustment or temporarily interruption by system organ class and preferred term during re-treatment phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the re-treatment phase | .358 |
| Table 14.3.1-6.3.2 Treatment-emergent adverse events occurrence requiring dosage adjustment or temporarily interruption by system organ class and preferred | |

| term during re-treatment phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the re-treatment phase | |
|---|---|
| Table 14.3.1-6.4.1 Treatment-emergent adverse events of interest incidence, regardless of study drug relationship, by specific group and preferred term during Pre-randomization Induction/consolidation phase –by treatment arm, overall and maximum grade 3/4 – Full Analysis Set | 359 |
| Table 14.3.1-6.4.2 Treatment-emergent adverse events of interest occurrence, regardless of study drug relationship, by specific group and preferred term during Pre-randomization Induction/consolidation phase – by treatment arm, overall and maximum grade 3/4 –Full Analysis Set | 360 |
| Table 14.3.1-6.5.1 Treatment-emergent adverse events of interest incidence by specific group and preferred term during post-randomization consolidation phase (ARM 2) – overall and maximum grade 3/4 – Subset of Full Analysis Set randomized to Arm 2 | 361 |
| Table 14.3.1-6.5.2 Treatment-emergent adverse events of interest occurrence, by specific group and preferred term during post-randomization consolidation phase (ARM 2) – overall and maximum grade 3/4 – Subset of Full Analysis Set randomized to Arm 2 | 362 |
| Table 14.3.1-6.6.1 Treatment-emergent adverse events of interest incidence by specific group and preferred term during re-treatment phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the re-treatment phase | 363 |
| Table 14.3.1-6.6.2 Treatment-emergent adverse events of interest occurrence by specific group and preferred term during re-treatment phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the re-treatment phase | |
| Table 14.3.1-6.7.1 Adverse events of interest incidence by specific group and preferred term during TFR phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the TFR phase | |
| Table 14.3.1-6.7.2 Adverse events of interest occurrence by specific group and preferred term during TFR phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the TFR phase | |
| Table 14.3.1-7.1.1 Treatment Emergent adverse events of interest incidence, regardless of study drug relationship, by specific group and preferred term and by cardiovascular risk factors during Pre-randomization Induction/consolidation phase – by treatment arm, overall and maximum grade 3/4 – Full Analysis Set | 365 |
| Table 14.3.1-7.1.2 Treatment Emergent adverse events of interest occurrence, regardless of study drug relationship, by specific group and preferred term and by cardiovascular risk factors during Pre-randomization Induction/consolidation phase – by treatment arm, overall and maximum grade 3/4 –Full Analysis Set | 366 |
| Table 14.3.1-7.2.1 Treatment-emergent adverse events of interest incidence, regardless of study drug relationship, during post-randomization consolidation phase (ARM 2), by specific group and preferred term, and by cardiovascular risk factor—overall and maximum grade 3 or 4 – Subset of Full Analysis Set randomized to Arm 2 | 367 |

| Table 14.3.1-7.2.2 Treatment-emergent adverse events of interest occurrence, regardless of study drug relationship, during post-randomization consolidation phase (ARM 2), by specific group and preferred term, and by cardiovascular risk factor – overall and maximum grade 3 or 4 – Subset of Full Analysis Set randomized to Arm 2 | .368 |
|---|---|
| Table 14.3.1-7.3.1 Treatment-emergent adverse events of interest incidence, regardless of study drug relationship, during re-treatment phase, by specific group and preferred term, and by cardiovascular risk factor – Subset of Full | .369 |
| Table 14.3.1-7.3.2 Treatment-emergent adverse events of interest occurrence, regardless of study drug relationship, during re-treatment phase, by specific group and preferred term, and by cardiovascular risk factor – Subset of Full Analysis Set entering the re-treatment phase. | .370 |
| Table 14.3.1-7.4.1 Adverse events of interest incidence, regardless of study drug relationship, during TFR phase, by specific group and preferred term, and by cardiovascular risk factor – Subset of Full Analysis Set entering the TFR phase | .371 |
| Table 14.3.1-7.4.2 Adverse events of interest occurrence, regardless of study drug relationship, during TFR phase, by specific group and preferred term, and by cardiovascular risk factor – Subset of Full Analysis Set entering the TFR phase | .371 |
| Table 14.3.1-7.5.1 Treatment-emergent adverse events of interest incidence, regardless of study drug relationship, during pre-randomization Induction/consolidation phase, by specific group and preferred term and by 4 cardiovascular risk factors – overall and maximum grade 3/4 –Full Analysis Set | |
| Table 14.3.1-7.5.2 Treatment-emergent adverse events of interest occurence, regardless of study drug relationship, during pre-randomization Induction/consolidation phase, by specific group and preferred term and by 4 cardiovascular risk factors – overall and maximum grade 3/4 –Full Analysis Set | 372 |
| Table 14.3.1-7.6.1 Treatment-emergent adverse events of interest incidence, regardless of study drug relationship, during post-randomization consolidation phase (ARM 2), by specific group and preferred term, and by 4 categories of cardiovascular risk factors— overall and maximum grade 3 or 4—Subset of Full Analysis Set randomized to Arm 2 | |
| Table 14.3.1-7.6.2 Treatment-emergent adverse events of interest occurrence, regardless of study drug relationship, during post-randomization consolidation phase (ARM 2), by specific group and preferred term, and by 4 categories of cardiovascular risk factors – overall and maximum grade 3 or 4 – Subset of Full Analysis Set randomized to Arm 2 | .372 |
| Table 14.3.1-7.7.1 Treatment-emergent adverse events of interest incidence, regardless of study drug relationship, during re-treatment phase, by specific group and preferred term, and by 4 categories of cardiovascular risk factors – Subset of Full Analysis Set entering the re-treatment phase | .373 |
| Table 14.3.1-7.7.2 Treatment-emergent adverse events of interest occurrence, regardless of study drug relationship, during re-treatment phase, by specific | |

| group and preferred term, and by 4 categories of cardiovascular risk factors—Subset of Full Analysis Set entering the re-treatment phase | .373 |
|---|---|
| Table 14.3.1-7.8.1 Adverse events of interest incidence, regardless of study drug relationship, during TFR phase, by specific group and preferred term, and by 4 categories of cardiovascular risk factors – Subset of Full Analysis Set entering the TFR phase | .374 |
| Table 14.3.1-7.8.2 Adverse events of interest occurrence, regardless of study drug relationship, during TFR phase, by specific group and preferred term, and by 4 categories of cardiovascular risk factors—Subset of Full Analysis Set entering the TFR phase | .374 |
| Table 14.3.1-9.1 On treatment deaths, by system organ class and preferred term during pre-randomization Induction/Consolidation phase - Safety Set | .375 |
| Table 14.3.1-9.2 On treatment deaths, by system organ class and preferred term during post-randomization consolidation phase (ARM 2) – Subset of Safety Set randomized to Arm 2 | .376 |
| Table 14.3.1-9.3 On treatment deaths, by system organ class and preferred term during re-treatment phase – Subset of Safety Set entering the re-treatment phase | .376 |
| Table 14.3.1-10.1.1 Cardiac and vascular adverse events of interest, incidence, by treatment arm during the pre-randomization induction/consolidation phase - | .377 |
| Table 14.3.1-10.1.2 Cardiac and vascular adverse events of interest, occurence, by treatment arm during the pre-randomization induction/consolidation phase - Full Analysis Set | .379 |
| Table 14.3.1-10.2.1 Cardiac and vascular adverse events of interest incidence, during the post-randomization consolidation phase (ARM 2) - Subset of Full Analysis Set randomized to Arm 2 | .380 |
| Table 14.3.1-10.2.2 Cardiac and vascular adverse events of interest occurrence, during the post-randomization consolidation phase (ARM 2) - Subset of Full Analysis Set randomized to Arm 2 | .381 |
| Table 14.3.1-10.3.1 Cardiac and vascular adverse events of interest, incidence, by treatment arm during the re-treatment phase – Subset of Full Analysis Set entered re-treatment phase | |
| Table 14.3.1-10.3.2 Cardiac and vascular adverse events of interest, occurence, by treatment arm during the re-treatment phase - Subset of Full Analysis Set entered re-treatment phase | .382 |
| Table 14.3.1-10.4.1 Cardiac and vascular adverse events of interest, incidence, by treatment arm during the TFR phase – Subset of Full Analysis Set entered TFR phase | .383 |
| Table 14.3.1-10.4.2 Cardiac and vascular adverse events of interest, occurence, by treatment arm during the TFR phase - Subset of Full Analysis Set entered TFR phase - | .383 |
| Table 14.3.1-10.5 Relationship between cardiac and vascular adverse events of interest with total cholesterol values - Full Analysis Set | .384 |
| Table 14.3.1-10.6 Relationship between cardiac and vascular adverse events of interest with glycemic values - Full Analysis Set | 385 |

| Table 14.3.1-11.1.1 Kaplan-Meier estimate of time-to-first CVEs during the pre-<br>randomization induction/consolidation phase – Full analysis set | 386 |
|---|---|
| Table 14.3.1-11.1.2 Kaplan-Meier estimate of time-to-first CVEs during the post-randomization consolidation phase (ARM 2)— Subset of Full Analysis Set | .389 |
| Table 14.3.1-11.2 Kaplan-Meier estimate of time-to-first CVEs during the retreatment phase – Subset of Full Analysis Set entering the re-treatment phase | 390 |
| Table 14.3.1-12.1 Medical history by system organ class and preferred term- Full Analysis Set | 391 |
| Table 14.3.1-13.1 Prior exposure to imatinib before screening, MMR, age, and Sokal by LSC detection category - LSC sub-study Full Analysis Set | 392 |
| Table 14.3.1-13.2.1 Percentage from total CD34+ cells, CD34+/CD38+ cells - Subgroup of LSC sub-study Full Analysis Set, LSC detected | .393 |
| Table 14.3.1-13.2.2 Percentage from total CD34+ cells, CD34+/CD38- cells - | 394 |
| Table 14.3.1-13.2.3 Percentage from total CD34+ cells, Immunophenotypically aberrant CD34+ cells - Subgroup of LSC sub-study Full Analysis Set, LSC detected | 394 |
| Table 14.3.1-13.2.4 Percentage from total CD34+ cells, Immunophenotypically aberrant CD34 negative cells - Subgroup of LSC sub-study Full Analysis Set, LSC detected | .395 |
| Table 14.3.1-13.3.1 Percentage of Ph+ cells, CD34+/CD38- cells - Subgroup of LSC sub-study Full Analysis Set, LSC detected | 395 |
| Table 14.3.1-13.3.2 Percentage of Ph+ cells, CD34+/CD38- cells - Subgroup of LSC sub-study Full Analysis Set, LSC detected | .395 |
| Table 14.3.1-13.3.3 Percentage of Ph+ cells, Immunophenotypically aberrant CD34+ cells - Subgroup of LSC sub-study Full Analysis Set, LSC detected | 395 |
| Table 14.3.1-13.3.4 Percentage of Ph+ cells, Immunophenotypically aberrant CD34 negative cells - Subgroup of LSC sub-study Full Analysis Set, LSC detected | 395 |
| Table 14.3.1-13.4 Total Percentage of CD34+ cells- Subgroup of LSC sub-study Full Analysis Set, LSC detected | .395 |
| Table 14.3.1-13.5 LSC detection - LSC sub-study Full Analysis Set | 396 |
| Section 14.3.2 – Listings of deaths, other serious and significant adverse events | 397 |
| Listing 14.3.2-1.1 Listing of deaths – Full Analysis Set | 397 |
| Listing 14.3.2-1.2 Listing of deaths SDV sensitivity – Full Analysis Set | 397 |
| Listing 14.3.2-2.1 Listing of adverse events of special interest – Full Analysis Set | 398 |
| Listing 14.3.2-2.2 Listing of adverse events leading to study drug discontinuation – Full Analysis Set | 398 |
| Listing 14.3.2-2.3 Listing of adverse events leading to study drug discontinuation during re-treatment phase – Subset of Full Analysis Set entering the retreatment period | 399 |
| Section 14.3.3 – Narratives of deaths, other serious and significant adverse events (non statistics and programming deliverables) | |
| Section 14.3.4 – Abnormal laboratory value listings | |
| $\sim$ | |

| Listing 14.3.4-1.1 Listing of abnormal hematology laboratory value – Full Analysis Set | 400 |
|---|---|
| Listing 14.3.4-2.1 Listing of abnormal biochemistry laboratory value – Full Analysis Set | |
| Section 16 – Appendices | 401 |
| Section 16.1 – Study information | 401 |
| Section 16.1.6 – Listing of patients receiving test drug(s)/investigational product(s) from specific batches where more than one batch was used | .401 |
| Section 16.1.7 – Randomization scheme and codes (subject identification and treatment assigned) | |
| Listing 16.1.7-1.1 Randomization schemes - Randomized patients | 402 |
| Section 16.1.9 – Documentation of statistical methods | 403 |
| Listing 16.1.9.1 Raw Statistical output from Demographic and characteristics at baseline– Full Analysis Set | .404 |
| Listing 16.1.9.1.1 Raw Statistical output from Demographic and characteristics at baseline– LSC sub-study Full Analysis Set | .404 |
| Listing 16.1.9.2 Raw Statistical output from History of prior Imatinib therapy – Full Analysis Set | .404 |
| Listing 16.1.9.2.1 Raw Statistical output from History of prior Imatinib therapy – LSC sub-study Full Analysis Set | .404 |
| Listing 16.1.9.3 Raw Statistical output from Cardiovascular risk factors at baseline – Full Analysis Set | .405 |
| Listing 16.1.9.4.1 Raw Statistical output from Molecular response MR4.0 at 12 months of TFR–Subset of Full Analysis Set entering the TFR phase | .405 |
| Listing 16.1.9.4.2 Raw Statistical output from Molecular response MR4.0 at 12 months of TFR-Subset of Per Protocol Analysis Set entering the TFR phase | .405 |
| Listing 16.1.9.5.1 Raw Statistical output from Kaplan-Meier analysis of treatment-free survival during the TFR phase – Subset of Full Analysis Set entering the TFR phase | .406 |
| Listing 16.1.9.5.2 Raw Statistical output from Kaplan-Meier analysis of treatment-free survival during the TFR phase – Subset of Per Protocol Analysis Set entering the TFR phase | .406 |
| Listing 16.1.9.5.3 Raw Statistical output from Kaplan-Meier analysis of overall survival from Randomization–Randomized Set | .406 |
| Listing 16.1.9.5.4 Raw Statistical output from Kaplan-Meier analysis of progression-free survival during the TFR phase – Subset of Full Analysis Set entering the TFR phase | .406 |
| Listing 16.1.9.6.1 Raw Statistical output from Kaplan-Meier estimate of time-to-first CVEs during the pre-randomization induction/consolidation phase – Full analysis set | .407 |
| Listing 16.1.9.6.2 Raw Statistical output from Kaplan-Meier estimate of time-to-<br>first CVEs during the post-randomization consolidation phase (ARM 2)—<br>Subset of Full Analysis Set nationts randomized on Arm 2 | 407 |
| annsecot fint Analysis aet natients fandomized on Afm / | 411/ |

| Listing 16.1.9.6.3 Raw Statistical output from Kaplan-Meier estimate of time-to-first CVEs during the re-treatment phase – Subset of Full Analysis Set entering the re-treatment phase | 407 |
|---|---|
| Section 16.2 – Patient data listings | |
| Listing 16.2-1.1 Enrolled patients | |
| Section 16.2.1 – Discontinued subjects | |
| Listing 16.2.1-1.1 Treatment and study completion - Safety Set | |
| Listing 16.2.1-1.2 Study discontinuation – Full Analysis Set | |
| Listing 16.2.1-1.3 Screen failures (All subjects enrolled) | |
| Section 16.2.2 – Protocol deviations | |
| Listing 16.2.2-1.1 Protocol deviations – Enrolled patients | |
| Section 16.2.3 – Patients excluded from the efficacy analysis | |
| Listing 16.2.3-1.1 Analysis set – All patients | |
| Section 16.2.4 – Demographics and data at screening | |
| Listing 16.2.4-1.1 Demographic data – Full Analysis Set | |
| Listing 16.2.4-2.1 Family history – Full Analysis Set | |
| Listing 16.2.4-2.2 Disease history– Full Analysis Set | 416 |
| Listing 16.2.4-3.1 Disease history I– Full Analysis Set | 417 |
| Listing 16.2.4-3.2 Disease history II– Full Analysis Set | 418 |
| Listing 16.2.4-3.3 Medical history/current medical condition – Full Analysis Set | 418 |
| Listing 16.2.4.4 Cardiovascular risk factors at baseline for patients with not evaluable CV risk factor, Full Analysis Set | 419 |
| Section 16.2.5 – Compliance and/or drug concentration data if available (including Bioanalytical Data Report) | 420 |
| Listing 16.2.5-1.1 Dosage administration records – Full Analysis Set | 420 |
| Section 16.2.6 – Individual efficacy response data | 420 |
| Listing 16.2.6-1.1 BCR-ABL(IS) ratio and molecular responses during Induction/Consolidation and post-randomization consolidation phase (ARM 2) – Full Analysis Set | 420 |
| Listing 16.2.6-1.2 BCR-ABL(IS) ratio and molecular responses during TFR phase – Subset of Full Analysis Set entering the TFR phase | |
| Listing 16.2.6-1.3 BCR-ABL(IS) ratio and molecular responses during re-treatment phase – Subset of Full Analysis Set entering the re-treatment phase | |
| Listing 16.2.6-2.1 Criteria of successful TFR – Subset of Full Analysis Set entering the TFR phase | 422 |
| Listing 16.2.6-3.1 Assessment of progression-free survival during the TFR phase – Subset of Full Analysis Set entering the TFR phase | 423 |
| Listing 16.2.6-3.2 Assessment of treatment-free survival during the TFR phase – Subset of Full Analysis Set entering the TFR phase | 424 |
| Listing 16.2.6-3.3 Assessment of overall survival From Randomization – Randomized set | 425 |

| Listing 16.2.6-3.4 Assessment of relapse and treatment status during the TFR phase —Subset of Full Analysis Set entering the TFR phase and relapsed | 426 |
|---|---|
| Listing 16.2.6-4.1 WBC and molecular response in patients with WBC increase | .427 |
| , | |
| Listing 16.2.6-5.1 Individual Efficacy data, Molecular response – Full Analysis Set | |
| Listing 16.2.6-5.2 Individual Efficacy data, Bone-marrow I – Full Analysis Set | |
| Listing 16.2.6-5.3 Individual Efficacy data, Bone -marrow II – Full Analysis Set | 430 |
| Listing 16.2.6-6.1.1 Total percentage of CD34+ cells – LSC sub-study Full Analysis Set | 431 |
| Listing 16.2.6-6.2.1 Percentage of cells from total CD34 positive— LSC sub-study Full Analysis Set | 432 |
| Listing 16.2.6-6.3.1 Number of events sorted– LSC sub-study Full Analysis Set | 433 |
| Listing 16.2.6-6.4.1 Ph+ by HIS- LSC sub-study Full Analysis Set | 434 |
| Listing 16.2.6-6.5.1 BCR-ABL by RT-PCR-LSC sub-study Full Analysis Set | 435 |
| Section 16.2.7 – Adverse event listings | 436 |
| Listing 16.2.7-1.1 All adverse events – Full Analysis Set | |
| Listing 16.2.7-2.1 Serious adverse events Full Analysis Set | |
| Listing 16.2.7-2.2 Adverse events leading to study drug discontinuation – Full Analysis Set | |
| Listing 16.2.7-2.3 Adverse events of interest – Full Analysis Set | |
| Listing 16.2.7-3.1 CV risk factors, Nilotinib exposure, glucose and total cholesterol rates for patients with cardiac and vascular adverse events of interest, Full | .440 |
| Listing 16.2.7-3.2 Cardiac and vascular adverse events of interest, Full Analysis Set | 441 |
| Listing 16.2.7-3.3 Outcomes and subsequent concomitant medications for patients with cardiac adverse events of interest, Full Analysis Set | .443 |
| Listing 16.2.7-3.4 Outcomes and subsequent concomitant medications for patients with vascular adverse events of interest, Full Analysis Set | 444 |
| · | |
| Listing 16.2.8-1.1 Hematology laboratory values and normal ranges – Full Analysis | .445 |
| | 443 |
| Listing 16.2.8-2.1 Biochemistry laboratory values and normal ranges – Full Analysis Set | 446 |
| Listing 16.2.8-3.1 Hematological data and molecular response in patients with absolute blasts higher than normal ranges, Full Analysis Set | 448 |
| Listing 16.2.8-3.2 Hematological data and molecular response in patients with absolute metamyelocytes higher than normal ranges, Full Analysis Set | 449 |
| Section 16.2.9 – Vital signs, physical findings and other observations related to | |
| safety listings | |
| Listing 16.2.9-1.1 Vital signs – Full Analysis Set | 450 |
| Listing 16.2.9-2.1 Electrocardiograms – Full Analysis Set | 451 |
| Listing 16.2.9-2.2 Echocardiography – Full Analysis Set | 451 |

| Listing 16.2.9-3.1 | Concomitant medications – Full Analysis Set | .452 |
|---|---|---|
| Listing 16.2.9- 3.2 | Prohibited concomitant medications – Full Analysis Set | .452 |
| Listing 16.2.9-4.1 | Prior Imatinib therapy– Full Analysis Set | .453 |
| Listing 16.2.9-4.2 | Prior antineoplastic therapy, other than Imatinib – Full Analysis | |
| Set | | .453 |
| Listing 16.2.9-5.1 | Survival follow-up- Full Analysis set | .454 |
| Listing 16.2.9-5.2 | Safety follow-up- Full Analysis set | .455 |
| Listing 16.2.9-6 I | Prior imatinib exposure – LSC sub-study Full Analysis Set | .456 |

# 1. General guidance

### 1.1 Document headers

The following header will be used for all tables, listings and figures in sections 14 and 16 outlined in this document: CAMN107AIC05.

## 1.2 Rules of presentation

Programming rules for tables and listings are described as follows.

- Add one space between a number and before the opening parenthesis and no spaces within the parenthesis e.g. 'xx (xx.x)' not 'xx(xx.x)'.
- There should be no spaces between a symbol and a number e.g. '<XX' and not '<XX'. A space is recommended between a special character and a number in order for a printout to print correctly, e.g. '≥ XX' instead of '≥XX'.
- There should be no '%' sign after a result in any data cell. The 'n (%)' should appear once in the column header or in the first column next to the variable name. If result = 0, then there should be no parenthesis with zero percentage only a zero e.g. '0' and not '0 (0.0)'. The same holds for estimates and their CIs when they are not estimable (NE), they should be presented as 'NE' and not 'NE (NE, NE)'.
- Confidence intervals (CI) are provided in parenthesis, separated by a coma and a space after e.g. '(xx.x, xx.x)'.
- All categorical data will be summarized by frequencies and percentages. Where categorical data is missing, a 'Missing' row will be included at the bottom with frequencies also presented.
- Decimal places will be as follows:
  - o 3 decimal places for p-values; if p-value is less than 0.001, it will be displayed as <0.001.
  - o 1 decimal place more than the original data is recorded to for means, medians and percentiles.
  - o Two decimal places more for standard errors and standard deviations.
  - o The same precision for minimums and maximums.
  - o Frequency distribution: % has 1 decimal place.
  - Confidence intervals are given with the same number of decimal places as for the associated estimate.
  - o If percentage = 100, no decimal is required and no percentage will be displayed if the frequency count is zero.
- Default summary statistics for a continuous variable include n, mean, median, standard deviation, 25<sup>th</sup> and 75<sup>th</sup> percentiles. For CSR outputs min and max are optional and have only been displayed if needed.
- For all laboratory parameters, 'SI' unit is used.
- For AE tables, the preferred term will be sorted by descending frequency, unless indicated otherwise.
- All listings will be sorted by country, center, patient number and visit/ event date.

- Partial dates (day and/or month missing) will be listed as partial (not missing), unless
  the date has been imputed, in which case then the imputed date will be listed and flagged.
- AE listings: when AE end date is missing, i.e., AE continued at final examination, "continuing" should be listed as the AE end date in the listings.
- Day is relative to 'day 1' (defined above) and is calculated as: date of interest 'Day 1' date + 1. For visits/events occurring prior to Day 1 the '+1' will be excluded, so the day before Day 1 is Day -1.
- Variables in days will be converted to different time unit if necessary, using following conversion rule.
  - 1 month = 30.4375 days
  - year = 365.25 days

#### 1.3 Document headers

The following header will be considered as standard for all CSR tables, listings and figures outlined in this document:

```
CAMN107AIC05 - UNBLINDED - ANALYSIS CUT-OFF/ DBL DATE: DDMMMYYYY DRAFT/FINAL ...
Location/Program name - rundate
```

As the study is an open-label trial only one version of the tables, listings and figures will be produced.

## 1.4 Presentation of table numbering and titles within this document

In order to facilitate the inclusion of a table of contents for all output, the format of the number and title for each layout should be in the Novstyle format "Non-TOC Heading" and therefore does not exactly match the layout that is intended for the final deliverable.

In practice, the numbering and title for all outputs defined in this document will be of the following formats respectively:

Listing XX.X-X.X

Title Title Title Title Title

Population

## 1.5 Treatment group labels and ordering

The following treatment labels will be used for all tables, listings and figures in the order provided here:

- ARM 1: the nilotinib 24 months treatment arm
- ARM 2: the nilotinib 36 months treatment arm
- Randomized (ARM 1 + ARM 2)
- Not Randomized

# 1.6 Distribution logistics

- in-text tables/figures
- Post-text tables/figures/listings
- Appendix tables/figures/listings

| | | Listing Figures History – Changes compared to previous version of RAP module 7.1 | 2 |
|---|---|---|---|
| 1. | | al guidance | |
| | 1.1 | Document headers | |
| | 1.2 | Rules of presentation | 38 |
| | 1.3 | Document headers | 39 |
| | 1.4 | Presentation of table numbering and titles within this document | 40 |
| | 1.5 | Treatment group labels and ordering | 40 |
| | 1.6 | Distribution logistics | 40 |
| 2. | Overa | ll table of contents for statistics and programming output | 41 |
| Tal | oles, Lis | sting Figures | 41 |
| 3. | Shells | and specification for CSR | 75 |
| | 3.1 | Shells and specifications for sections 10 of the CSR (In-textText tables, listings and figures) | 75 |
| | Sectio | n 10 | 109 |
| | Table | 10-1 Analysis sets – All patients | 109 |
| | Table | 10-2 Patient disposition during Induction/Consolidation phase and post-Randomization Consolidation phase -Enrolled patients | 110 |
| | Table | 10-3 Demographic and characteristics at baseline – Full Analysis Set | 111 |
| | Table | 10-4 Disease history – Full Analysis Set. | 113 |
| | Table | 10-5 Duration of exposure to study treatment during pre-randomization Induction/Consolidation Safety Set | 116 |
| | Table | 10-6 Duration of exposure to study treatment during post-randomization Consolidation phase (ARM 2) - Subset of Safety Set randomized to Arm 2 | 116 |
| | Table | 11-1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase – Full Analysis Set | 117 |
| | Table | 11-2 Raw cumulative incidence of MR 4.0 during post-randomization consolidation phase (ARM 2) - Subset of Full Analysis Set randomized to Arm 2 | 117 |
| | Table | 11-3 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase – Full Analysis Set | 117 |
| | Table | 11-4 Raw cumulative incidence of MR 4.5 during post-randomization consolidation phase (ARM 2) - Subset of Full Analysis Set randomized to Arm 2 | 118 |
| | Table | 11-5 Primary endpoint, Molecular response MR4.0 at 12 months of TFR phase—Subset of Full Analysis Set entering the TFR phase | 118 |
| | Table | 11-6 Secondary endpoint Kaplan-Meier analysis of treatment-free survival during the TFR phase – Subset of Full Analysis Set entering the TFR phase | 119 |
| | Table | 11-7 Secondary endpoint, Molecular response 4.0 during post-randomization consolidation phase (ARM 2) – Subset of Full Analysis Set randomized to Arm 2 | 120 |

| Table 11-8 Secondary endpoint, Kaplan-Meier analysis of overall survival from Randomization–Randomized Set | 21 |
|---|---|
| Table 12-1 Overall summary of treatment-emergent adverse events occurring during pre-randomization Induction/consolidation phase – Full Analysis Set | 22 |
| Table 12-2 Overall summary of treatment-emergent adverse events occurring during post-randomization consolidation phase (ARM 2) – Subset of Full Analysis Set randomized to Arm 2 | 23 |
| Table 12-3 Overall summary of treatment-emergent adverse events occurring during re-treatment phase – Subset of Full Analysis Set entering the re-treatment phase | 24 |
| Table 12-4 Overall summary of adverse events occurring during TFR phase – Subset of Full Analysis Set entering the TFR phase | 25 |
| Table 12-5 Overall summary of frequent [1] treatment-emergent adverse events occurring during pre-randomization Induction/consolidation phase – Full Analysis Set | 26 |
| Table 12-6 Overall summary of frequent [1] treatment-emergent adverse events occurring during post-randomization Consolidation phase (ARM 2) – Subset of Full Analysis Set randomized to Arm 2 | 26 |
| Table 12-7 Overall summary of frequent [1] treatment-emergent adverse events occurring during re-treatment phase – Subset of Full Analysis Set entering the re-treatment phase — 12 | 26 |
| Table 12-8 Overall summary of frequent [1] adverse events occurring during TFR phase – Subset of Full Analysis Set entering the TFR phase | 26 |
| Table 12-9 Serious treatment-emergent adverse events incidence, regardless of study drug relationship, by system organ class and preferred term during prerandomization Induction/consolidation phase – overall and maximum grade 3/4 –Full Analysis Set | 27 |
| Table 12-10 Serious treatment-emergent adverse events incidence, regardless of study drug relationship, by system organ class and preferred term during post-randomization consolidation phase (ARM 2) – overall and maximum grade 3/4 – Subset of Full Analysis Set randomized to Arm 2 | 28 |
| Table 12-11 Serious treatment-emergent adverse events incidence, regardless of study drug relationship, by system organ class and preferred term during retreatment phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the re-treatment phase | 28 |
| Table 12-12 Serious adverse events incidence, regardless of study drug relationship, by system organ class and preferred term during TFR phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the TFR phase 12 | 28 |
| Table 12-13 Treatment-emergent adverse events of interest incidence, regardless of study drug relationship, by specific group and preferred term during Prerandomization Induction/consolidation phase –by treatment arm, overall and maximum grade 3/4 – Full Analysis Set | |
| Table 12-14 Treatment-emergent adverse events of interest incidence by specific group and preferred term during post-randomization Consolidation phase (ARM 2) – overall and maximum grade 3/4 – Subset of Full Analysis Set randomized to Arm 2. | 30 |

| Table 12-15 Treatment-emergent adverse events of interest incidence by specific group and preferred term during re-treatment phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the re-treatment phase | 131 |
|---|---|
| Table 12-16 Adverse events of interest incidence by specific group and preferred term during TFR phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the TFR phase | 131 |
| Table 12-17 Treatment-emergent adverse events incidence leading to study drug discontinuation by system organ class and preferred term during prerandomization Induction/Consolidation phase – overall and maximum grade 3/4 –Full Analysis Set | 132 |
| Table 12-18 Treatment-emergent adverse events incidence leading to study drug discontinuation by system organ class and preferred term during post-randomizationphase (ARM 2) – overall and maximum grade 3/4 – Subset of Full Analysis Set randomized to Arm 2 | 133 |
| Table 12-19 On treatment deaths, by system organ class and preferred term during pre-randomization Induction/Consolidation phase - Safety Set | 133 |
| Table 12-20 On treatment deaths, by system organ class and preferred term during post-randomization consolidation phase (ARM 2) – Subset of Safety Set randomized to Arm 2 | 134 |
| Table 12-21 On treatment deaths, by system organ class and preferred term during re-treatment phase – Subset of Safety Set entering the re-treatment phase | 134 |
| Listing 12-1 Listing of deaths – Full Analysis Set | 135 |
| Figure 11-1 Primary endpoint, Bar plot MR4.0 at 12 months of TFR phase –Subset of Full Analysis Set entering the TFR phase | 136 |
| Figure 11-2 Kaplan-Meier analysis of treatment-free survival during the TFR phase —Subset of Full Analysis Set entering the TFR phase | 137 |
| 3.2 Shells and specifications for Sections 14 and 16 of the CSR | 138 |
| Section 14 – tables, figures and graphs referred to but not included in the text | 138 |
| Section 14.1 – Demographic data | 138 |
| Table 14.1-1.1 Enrollment by country and center – All patients | 139 |
| Table 14.1-1.2 Randomization by country and center – Randomized patients | 140 |
| Table 14.1-1.3 Patient disposition (Screening failures), All patients | 141 |
| Table 14.1-2.1 Patient disposition during Induction/Consolidation phase and post-Randomization Consolidation phase -Enrolled patients | 143 |
| Table 14.1-2.2 Patient disposition in each randomized arm – Full Analysis Set | 144 |
| Table 14.1-2.2.1 Patient disposition – Enrolled patients in LSC substudy | 147 |
| Table 14.1-2.3 Analysis sets –All patients | 148 |
| Table 14.1-2.4 Not Randomized patients - Enrolled patients | 149 |
| Table 14.1-2.5 Patient disposition, Overall and by year-phase -Enrolled patients | 150 |
| Table 14.1-2.6 Patients discontinued and reason for discontinuation – Full Analysis Set | 154 |
| Table 14.1-2.6.1 Patients discontinued and reason for discontinuation, SDV | |
| sensitivity – Full Analysis Set | 156 |

| Table 14.1-2.7 Summary of TFR phase – Full Analysis Set | .157 |
|---|---|
| Table 14.1-2.7.1 Summary of TFR phase, SDV sensitivity – Full Analysis Set | |
| Table 14.1-2.8 Summary of re-treatment phase – Full Analysis Set | .159 |
| Table 14.1-2.8.1 Summary of re-treatment phase, SDV sensitivity – Full Analysis Set | .160 |
| Table 14.1-2.9 Summary of patients with relapse during the TFR phase but no entering re-treatment phase —Subset of Full Analysis Set entering the TFR phase | 161 |
| Table 14.1-3.1 Demographic and characteristics at baseline– Full Analysis Set | |
| Table 14.1-3.1.1 Demographic and characteristics at baseline– LSC sub-study Full Analysis Set | |
| Table 14.1-4.1 Disease history – Full Analysis Set | |
| Table 14.1-4.1.1 Disease history – LSC sub-study Full Analysis Set | |
| Table 14.1-5.1 History of prior Imatinib therapy – Full Analysis Set | |
| Table 14.1-5.1.1 History of prior Imatinib therapy – LSC sub-study Full Analysis Set. | |
| Table 14.1-5.2 Prior antineoplastic therapy, other than Imatinib, by ATC class and preferred term - Full Analysis Set | |
| Table 14.1-6.1 Cardiovascular risk factors at baseline – Full Analysis Set | |
| Table 14.1-6.2 Cardiovascular risk factors (based on medical history, laboratory | . 1 / 1 |
| values and vital signs at baseline) – Full Analysis Set | .175 |
| Section 14.2 – Efficacy and other non-safety data (e.g. PK, PK/PD, Health Econ., QoL) | .177 |
| Figure 14.2-1.1 Box-plot of BCR-ABL ratio (IS) during pre-randomization Induction/Consolidation phase – Full Analysis Set | .178 |
| Figure 14.2-1.2 Box-plot of BCR-ABL ratio (IS) during post-randomization<br>Consolidation phase (ARM 2) – Subset of Full Analysis Set randomized to<br>ARM 2 | .179 |
| Figure 14.2-1.3 Box-plot of BCR-ABL ratio (IS) during TFR phase – Subset of Full Analysis Set entered TFR | .179 |
| Figure 14.2-1.4 Box-plot of BCR-ABL ratio (IS) during re-treatment phase – Subset of Full Analysis Set entered re-treatment | .179 |
| Figure 14.2-1.5 Box-plot of BCR-ABL ratio (IS) during TFR phase – , SDV sensitivity Subset of Full Analysis Set entered TFR | .180 |
| Figure 14.2-1.6 Box-plot of BCR-ABL ratio (IS) during re-treatment phase, SDV sensitivity –Subset of Full Analysis Set entered re-treatment | .180 |
| Figure 14.2-2.1.1 Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase - Full Analysis Set | .181 |
| Figure 14.2-2.1.2 Raw cumulative incidence of MMR during post-randomization Consolidation phase (ARM 2) - Subset of Full Analysis Set randomized to ARM 2 | .181 |
| Figure 14.2-2.2.1 Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase by halving time of BCR-ABL (IS) ratio - Full Analysis Set | 182 |

| Figure | 14.2-2.2.2 Raw cumulative incidence of MMR during post-randomization Consolidation phase (ARM 2) by halving time of BCR-ABL (IS) ratio - Subset of Full Analysis Set randomized to ARM 2 | 182 |
|---|---|---|
| Figure | 14.2-2.3.1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase – Full Analysis Set | 183 |
| Figure | 14.2-2.3.2 Raw cumulative incidence of MR 4.0 during post-randomization Consolidation phase (ARM 2) - Subset of Full Analysis Set randomized to ARM 2 | 183 |
| Figure | 14.2-2.3.11 Raw cumulative incidence of MR 4.0, Randomized vs Not Randomized, during pre-randomization Induction/Consolidation phase - Full Analysis Set | 184 |
| Figure | 14.2-2.4.1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase by halving time of BCR-ABL (IS) ratio - Full Analysis Set | 184 |
| Figure | 14.2-2.4.2 Raw cumulative incidence of MR 4.0 during post-randomization Consolidation phase (ARM 2) by halving time of BCR-ABL (IS) ratio - Subset of Full Analysis Set randomized to ARM 2 | 185 |
| Figure | 14.2-2.5.1 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase - Full Analysis Set | 185 |
| Figure | 14.2-2.5.11 Raw cumulative incidence of MR 4.5, Randomized vs Not Randomized, during pre-randomization Induction/Consolidation phase-Full Analysis Set | 185 |
| Figure | 14.2-2.5.2 Raw cumulative incidence of MR 4.5 during post-randomization Consolidation phase (ARM 2) - Subset of Full Analysis Set randomized to ARM 2 | 185 |
| Figure | 14.2-2.6.1 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase by halving time of BCR-ABL (IS) ratio - Full Analysis Set | 185 |
| Figure | 14.2-2.6.2 Raw cumulative incidence of MR 4.5 during post-randomization Consolidation phase (ARM 2) by halving time of BCR-ABL (IS) ratio - Subset of Full Analysis Set randomized to ARM 2 | 186 |
| Figure | 14.2-2.7.1 Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase - Full Analysis Set patients not reaching MMR at baseline | 186 |
| Figure | 14.2-2.8.1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase - Full Analysis Set patients not reaching MR 4.0 at baseline | |
| Figure | 14.2-2.9.1 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase - Full Analysis Set patients not reaching MR 4.5 at baseline | |
| Figure | 14.2-2.9.2 Raw cumulative incidence of MR 4.5 during post-randomization Induction/Consolidation phase (ARM 2)- Subset of Full Analysis Set patients not reaching MR 4.5 at baseline, randomized to ARM 2 | 186 |
| Figure | 14.2-2.10.1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase by BCR-ABL(IS) ratio at baseline - Full | 187 |

| Figure 14.2-2.10.2 Raw cumulative incidence of MR 4.0 during post-randomization Consolidation phase (ARM 2) by BCR-ABL(IS) ratio at baseline - Subset of Full Analysis Set randomized to ARM 2 |
|---|
| Figure 14.2-2.11.1 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase by BCR-ABL(IS) ratio at baseline - Full Analysis Set |
| Figure 14.2-2.11.2 Raw cumulative incidence of MR 4.5 during post-randomization Consolidation phase (ARM 2) by BCR-ABL(IS) ratio at baseline - Subset of Full Analysis Set randomized to ARM 2 |
| Figure 14.2-2.12.1 Box-plot of BCR-ABL ratio (IS) during pre-randomization Induction/Consolidation phase, excluding outliers (BCR-ABL (IS) ratio>10 - Full Analysis Set |
| Figure 14.2-2.12.2 Box-plot of BCR-ABL ratio (IS) over post-randomization Consolidation phase (ARM 2), excluding outliers (BCR-ABL (IS) ratio>10 - Subset of Full Analysis Set randomized to ARM 2 |
| Figure 14.2-13.1 Raw cumulative incidence of loss of MMR during TFR – Subset of Full Analysis Set entering the TFR phase |
| Figure 14.2-13.2 Raw cumulative incidence of MMR during re-treatment phase – Subset of Full Analysis Set entering the re-treatment phase |
| Figure 14.2-13.3 Raw cumulative incidence of loss of MMR during TFR, SDV sensitivity – Subset of Full Analysis Set entering the TFR phase |
| Figure 14.2-13.4 Raw cumulative incidence of MMR during re-treatment phase, SDV sensitivity – Subset of Full Analysis Set entering the re-treatment phase. 192 |
| Figure 14.2-14.1 Raw cumulative incidence of loss of MR4.0 during TFR phase – Subset of Full Analysis Set entering the TFR phase |
| Figure 14.2-14.2 Raw cumulative incidence of MR4.0 during re-treatment phase – Subset of Full Analysis Set entering the re-treatment phase |
| Figure 14.2-14.3 Raw cumulative incidence of loss of MR4.0 during TFR phase, SDV sensitivity –Subset of Full Analysis Set entering the TFR phase193 |
| Figure 14.2-14.4 Raw cumulative incidence of MR4.0 during re-treatment phase, SDV sensitivity – Subset of Full Analysis Set entering the re-treatment phase 193 |
| Figure 14.2-15.1 Raw cumulative incidence of loss of MR4.5 during TFR phase – Subset of Full Analysis Set entering the TFR phase with MR4.5 |
| Figure 14.2-15.2 Raw cumulative incidence of MR4.5 during re-treatment phase – Subset of Full Analysis Set entering the re-treatment phase |
| Figure 14.2-15.3 Raw cumulative incidence of loss of MR4.5 during TFR phase, SDV sensitivity – Subset of Full Analysis Set entering the TFR phase with MR4.5 |
| Figure 14.2-15.4 Raw cumulative incidence of MR4.5 during re-treatment phase, SDV sensitivity – Subset of Full Analysis Set entering the re-treatment phase 194 |
| Figure 14.2-16 Bar plot MR4.0 at 12 months of TFR phase –Subset of Full Analysis Set entering the TFR phase |
| Figure 14.2-16.2 Bar plot MR4.0 at month 12 TFR phase, SDV sensitivity –Subset of Full Analysis Set entering the TFR phase |

| Figure 14.2-17.1 Kaplan-Meier analysis of progression-free survival during the TFR phase –Subset of Full Analysis Set entering the TFR phase | 96 |
|---|---|
| Figure 14.2-17.2 Kaplan-Meier analysis of treatment-free survival during the TFR phase –Subset of Full Analysis Set entering the TFR phase | 96 |
| Figure 14.2-17.3 Kaplan-Meier analysis of progression-free survival during the TFR phase, SDV sensitivity –Subset of Full Analysis Set entering the TFR phase 19 | <del>9</del> 7 |
| Figure 14.2-17.4 Kaplan-Meier analysis of treatment-free survival during the TFR phase, SDV sensitivity –Subset of Full Analysis Set entering the TFR phase 19 | <del>9</del> 7 |
| Figure 14.2-18.1 Kaplan-Meier analysis of reachievement of MMR, after loss of response in TFR –Subset of Full Analysis Set entering the re-treatment phase 19 | <del>9</del> 7 |
| Figure 14.2-18.2 Kaplan-Meier analysis of reachievement of MR4.0, after loss of response in TFR – Subset of Full Analysis Set entering the re-treatment phase. 19 | <b>97</b> |
| Figure 14.2-18.3 Kaplan-Meier analysis of reachievement of MMR, after loss of response in TFR, SDV sensitivity –Subset of Full Analysis Set entering the re-treatment phase | 98 |
| Figure 14.2-18.4 Kaplan-Meier analysis of reachievement of MR4.0, after loss of response in TFR, SDV sensitivity – Subset of Full Analysis Set entering the re-treatment phase | |
| Table 14.2-1.1 Description of BCR-ABL (IS) ratio at Month 3 and halving time of BCR-ABL (IS) ratio subgroups – Full Analysis Set | 99 |
| Table 14.2-2.1.1 Molecular response MR4.0 at 12 months of TFR–Subset of Full Analysis Set entering the TFR phase | 00 |
| Table 14.2-2.1.2 Molecular response MR4.0 at 12 months of TFR—Subset of Per Protocol Analysis Set entering the TFR phase | 00 |
| Table 14.2-2.1.3 Molecular response MR4.0 at 12 months of TFR–Full Analysis Set20 | )1 |
| Table 14.2-2.1.4 Molecular response MR4.0 at 12 months of TFR–Per Protocol Analysis Set | 01 |
| Table 14.2-2.1.5 Molecular response MR4.0 at 12 months of TFR—Subset of Full Analysis Set entering the TFR phase with MR4.0 achieved up to month 3 of pre-randomization Induction/Consolidation phase | 02 |
| Table 14.2-2.1.6 Molecular response MR4.0 at 12 months of TFR—Subset of Full Analysis Set entering the TFR phase with MR4.5 achieved up to month 3 of pre-randomization Induction/Consolidation phase | 02 |
| Table 14.2-2.1.7 Molecular response MR4.0 at 12 months of TFR, SDV sensitivity – Subset of Full Analysis Set entering the TFR phase | 02 |
| Table 14.2-2.1.8 Molecular response MR4.0 at 12 months of TFR, SDV sensitivity – Subset of Per Protocol Analysis Set entering the TFR phase20 | 02 |
| Table 14.2-2.1.9 Molecular response MR4.0 at 12 months of TFR, SDV sensitivity – Full Analysis Set | |
| Table 14.2-2.1.10 Molecular response MR4.0 at 12 months of TFR, SDV sensitivity —Per Protocol Analysis Set | |
| Table 14.2-2.2.1 Kaplan-Meier analysis of treatment-free survival during the TFR phase – Subset of Full Analysis Set entering the TFR phase20 | |

| Table 14.2-2.2.2 Kaplan-Meier analysis of treatment-free survival during the TFR phase – Subset of Per Protocol Analysis Set entering the TFR phase | 205 |
|---|---|
| Table 14.2-2.2.3 Kaplan-Meier analysis of treatment-free survival during the TFR phase, SDV sensitivity – Subset of Full Analysis Set entering the TFR phase. | 205 |
| Table 14.2-2.2.4 Kaplan-Meier analysis of treatment-free survival during the TFR phase, SDV sensitivity – Subset of Per Protocol Analysis Set entering the TFR phase | 205 |
| Table 14.2-2.3 Kaplan-Meier analysis of overall survival from Randomization— Randomized Set | 206 |
| Table 14.2-2.4 Kaplan-Meier analysis of progression-free survival during the TFR phase — Subset of Full Analysis Set entering the TFR phase | 207 |
| Table 14.2-2.5 Kaplan-Meier analysis of overall survival from Randomization, SDV sensitivity –Randomized Set | |
| Table 14.2-2.6 Kaplan-Meier analysis of progression-free survival during the TFR phase, SDV sensitivity — Subset of Full Analysis Set entering the TFR phase | .208 |
| Table 14.2-3.1 Major molecular response during pre-randomization Induction/Consolidation phase –Full Analysis Set | 209 |
| Table 14.2-3.1.1 Major molecular response during pre-randomization<br>Induction/Consolidation phase – LSC sub-study Full Analysis Set | 210 |
| Table 14.2-3.2 Major molecular response during post-randomization consolidation phase (ARM 2)— Subset of Full Analysis Set randomized to Arm 2 | 211 |
| Table 14.2-3.2.1 Major molecular response during post-randomization consolidation phase (ARM 2) – LSC sub-study Full Analysis Set randomized to Arm 2 | |
| Table 14.2-3.3 Major molecular response during TFR phase –Subset of Full Analysis Set patients entered TFR phase | |
| Table 14.2-3.4 Major molecular response during re-treatment phase–Subset of Full Analysis Set patients entered re- treatment phase | 213 |
| Table 14.2-3.5 Major molecular response during TFR phase –Subset of Full Analysis Set patients entered TFR phase with MR4.0 achieved up to month 3 of prerandomization Induction/Consolidation phase | |
| Table 14.2-3.6 Major molecular response during TFR phase –Subset of Full Analysis Set patients entered TFR phase with MR4.5 achieved up to month 3 of prerandomization Induction/Consolidation phase | |
| Table 14.2-3.7 Major molecular response during TFR phase, SDV sensitivity – Subset of Full Analysis Set patients entered TFR phase | 214 |
| Table 14.2-3.8 Major molecular response during re-treatment phase, SDV sensitivity —Subset of Full Analysis Set patients entered re- treatment phase | |
| Table 14.2-4.1 Molecular response 4.0 during pre-randomization Induction/Consolidation phase – Full Analysis Set | |
| Table 14.2-4.1.1 Molecular response 4.0 during pre-randomization Induction/Consolidation phase – LSC sub-study Full Analysis Set | |
| Table 14.2-4.2.1 Molecular response 4.0 during post-randomization consolidation phase (ARM 2) – Subset of Full Analysis Set randomized to Arm 2 | |

| Table 14.2-4.2.2 Molecular response 4.0 during post-randomization consolidation phase (ARM 2) – Subset of Per Protocol randomized to Arm 2 | 215 |
|---|---|
| Table 14.2-4.2.11 Molecular response 4.0 during post-randomization consolidation phase (ARM 2) – Subset of LSC sub-study Full Analysis Set randomized t Arm 2 | |
| Table 14.2-4.3.1 Molecular response 4.0 during TFR phase – Subset of Full Analysis Set entering the TFR phase | |
| Table 14.2-4.3.2 Molecular response 4.0 during TFR phase – Subset of Per Protoco Analysis Set entering the TFR phase | |
| Table 14.2-4.3.3 Molecular response 4.0 during TFR phase , SDV sensitivity – Subset of Full Analysis Set entering the TFR phase | 216 |
| Table 14.2-4.4 Molecular response 4.0 during re-treatment phase – Subset of Full Analysis Set entering the re-treatment phase | 217 |
| Table 14.2-4.5 Molecular response 4.0 during TFR phase – Subset of Full Analysis Set entering the TFR phase with MR4.0 achieved up to month 3 of prerandomization Induction/Consolidation phase | |
| Table 14.2-4.6 Molecular response 4.0 during TFR phase – Subset of Full Analysis Set entering the TFR phase with MR4.5 achieved up to month 3 of prerandomization Induction/Consolidation phase | |
| Table 14.2-4.7 Molecular response 4.0 during re-treatment phase, SDV sensitivity Subset of Full Analysis Set entering the re-treatment phase | |
| Table 14.2-5.1 Molecular response 4.5 during pre-randomization<br>Induction/Consolidation—Full Analysis Set | 218 |
| Table 14.2-5.1.1 Molecular response 4.5 during pre-randomization Induction/Consolidation— LSC sub-study Full Analysis Set | 218 |
| Table 14.2-5.2 Molecular response 4.5 during post-randomization consolidation phase (ARM 2) – Subset of Full Analysis Set randomized to Arm 2 | 218 |
| Table 14.2-5.2.1 Molecular response 4.5 during post-randomization consolidation phase (ARM 2) – Subset of LSC sub-study Full Analysis Set randomized to Arm 2 | |
| Table 14.2-5.3 Molecular response 4.5 during TFR phase – Subset of Full Analysis Set entering the TFR phase | S |
| Table 14.2-5.4 Molecular response 4.5 during re-treatment phase — Subset of Full Analysis Set entering the re-treatment phase | 218 |
| Table 14.2-5.5 Molecular response 4.5 during TFR phase – Subset of Full Analysis Set entering the TFR phase with MR4.0 achieved up to month 3 of prerandomization Induction/Consolidation phase | |
| Table 14.2-5.6 Molecular response 4.5 during TFR phase – Subset of Full Analysis Set entering the TFR phase with MR4.5 achieved up to month 3 of prerandomization Induction/Consolidation phase | |
| Table 14.2-5.7 Molecular response 4.5 during TFR phase, SDV sensitivity – Subse of Full Analysis Set entering the TFR phase | |
| Table 14.2-5.8 Molecular response 4.5 during re-treatment phase, SDV sensitivity Subset of Full Analysis Set entering the re-treatment phase | |

| Table 14.2-6.1 Raw cumulative incidence MMR during pre-randomization Induction/Consolidation phase – Full Analysis Set | 220 |
|---|---|
| Table 14.2-6.1.1 Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase – LSC sub-study Full Analysis Set | 221 |
| Table 14.2-6.2 Raw cumulative incidence MMR during post-randomization Consolidation phase (ARM 2) - Subset of Full Analysis Set patients randomized to ARM 2 | 221 |
| Table 14.2-6.2.1 Raw cumulative incidence MMR during post-randomization Consolidation phase (ARM 2) - Subset of LSC sub-study Fulls Anslysis Set randomized to ARM 2 | t<br>221 |
| Table 14.2-6.3 Raw cumulative incidence of MMR during re-treatment phase – Subset of Full Analysis Set entering the re-treatment phase | 222 |
| Table 14.2-6.4 Raw cumulative incidence of MMR during re-treatment phase , SDV sensitivity – Subset of Full Analysis Set entering the re-treatment phase | |
| Table 14.2-7.1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase – Full Analysis Set | 222 |
| Table 14.2-7.1.1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase – LSC sub-study Full Analysis Set | 222 |
| Table 14.2-7.2 Raw cumulative incidence of MR 4.0 during post-randomization consolidation phase (ARM 2) – Subset of Full Analysis Set randomized to ARM 2 | 223 |
| Table 14.2-7.2.1 Raw cumulative incidence of MR 4.0 during post-randomization consolidation phase (ARM 2) – Subset of LSC sub-study Full Analysis Set randomized to ARM 2 | 223 |
| Table 14.2-7.3 Raw cumulative incidence of MR 4.0 during re-treatment phase – Subset of Full Analysis Set entering the re-treatment phase | 223 |
| Table 14.2-7.4 Raw cumulative incidence of MR 4.0 during re-treatment phase, SDV sensitivity – Subset of Full Analysis Set entering the re-treatment phase | |
| Table 14.2-8.1 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase – Full Analysis Set | 224 |
| Table 14.2-8.1.1 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase – LSC sub-study Full Analysis Set | 224 |
| Table 14.2-8.2 Raw cumulative incidence of MR 4.5 during post-randomization consolidation phase (ARM 2) - Subset of Full Analysis Set randomized to Arm 2 | 224 |
| Table 14.2-8.2.1 Raw cumulative incidence of MR 4.5 during post-randomization consolidation phase (ARM 2) - Subset of LSC sub-study Full Analysis Set randomized to Arm 2 | 224 |
| Table 14.2-8.3 Raw cumulative incidence of MR 4.5 during re-treatment phase - Subset of Full Analysis Set entering the re-treatment phase | |
| Table 14.2-8.4 Raw cumulative incidence of MR 4.5 during re-treatment phase, SDV sensitivity - Subset of Full Analysis Set entering the re-treatment phase | |
| Table 14.2-9.1 Raw cumulative incidence of MMR during pre-randomization<br>Induction/Consolidation phase by halving time of BCR-ABL (IS) ratio – Full<br>Analysis Set | l<br>226 |

| Table 14.2-9.1.1 Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase by halving time of BCR-ABL (IS) ratio – LSC sub-study Full Analysis Set | .226 |
|---|---|
| Table 14.2-9.2 Raw cumulative incidence of MMR during post-randomization consolidation phase (ARM 2) by halving time of BCR-ABL (IS) ratio - Subset of Full Analysis Set randomized to Arm 2 | .227 |
| Table 14.2-9.2.1 Raw cumulative incidence of MMR during post-randomization consolidation phase (ARM 2) by halving time of BCR-ABL (IS) ratio - Subset of LSC sub-study Full Analysis Set randomized to Arm 2 | .228 |
| Table 14.2-9.3 Raw cumulative incidence of MMR during re-treatment phase by halving time of BCR-ABL (IS) ratio – Subset of Full Analysis Set entering the re-treatment phase | .228 |
| Table 14.2-10.1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase by halving time of BCR-ABL (IS) ratio – Full Analysis Set | .229 |
| Table 14.210.1.1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase by halving time of BCR-ABL (IS) ratio – LSC sub-study Full Analysis Set | .229 |
| Table 14.2-10.2 Raw cumulative incidence of MR 4.0 during post-randomization consolidation phase (ARM 2) by halving time of BCR-ABL (IS) ratio - Subset of Full Analysis Set randomized to Arm 2 | .229 |
| Table 14.2-10.2.1 Raw cumulative incidence of MR 4.0 during post-randomization consolidation phase (ARM 2) by halving time of BCR-ABL (IS) ratio - Subset of LSC sub-study Full Analysis Set randomized to Arm 2 | .229 |
| Table 14.2-10.3 Raw cumulative incidence of MR4.0 during re-treatment phase by halving time of BCR-ABL (IS) ratio – Subset of Full Analysis Set entering the re-treatment phase | .229 |
| Table 14.2-11.1 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase by halving time of BCR-ABL (IS) ratio – Full Analysis Set | .230 |
| Table 14.211.1.1 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase by halving time of BCR-ABL (IS) ratio – LSC sub-study Full Analysis Set | .230 |
| Table 14.2-11.2 Raw cumulative incidence of MR 4.5 during post-randomization consolidation phase (ARM 2) by halving time of BCR-ABL (IS) ratio - Subset of Full Analysis Set randomized to Arm 2 | .230 |
| Table14.2-11.2.1 Raw cumulative incidence of MR 4.5 during post-randomization consolidation phase (ARM 2) by halving time of BCR-ABL (IS) ratio - Subset of LSC sub-study Full Analysis Set randomized to Arm 2 | .230 |
| Table 14.2-11.3 Raw cumulative incidence of MR4.5 during re-treatment phase by halving time of BCR-ABL (IS) ratio – Subset of Full Analysis Set entering the re-treatment phase | |
| Table 14.2-12.1 Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase by BCR-ABL (IS) ratio at Month 3 – Full Analysis Set | 231 |

| Table 14.2-12.1.1 Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase by BCR-ABL (IS) ratio at Month 3 – LSC sub-study Full Analysis Set | 231 |
|---|---|
| Table 14.2-12.2 Raw cumulative incidence of MMR during post-randomization consolidation phase (ARM 2) by BCR-ABL (IS) ratio at Month 3 - Subset of Full Analysis Set randomized to Arm 2 | 231 |
| Table 14.2-12.2.1 Raw cumulative incidence of MMR during post-randomization consolidation phase (ARM 2) by BCR-ABL (IS) ratio at Month 3 - Subset of LSC sub-study Full Analysis Set randomized to Arm 2 | 232 |
| Table 14.2-12.3 Raw cumulative incidence of MMR during re-treatment phase by BCR-ABL (IS) ratio at Month 3 – Subset of Full Analysis Set entering the retreatment phase | 232 |
| Table 14.2-13.1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase by BCR-ABL (IS) ratio at Month 3 – Full Analysis Set | 233 |
| Table 14.2-13.1.1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase by BCR-ABL (IS) ratio at Month 3 – LSC sub-study Full Analysis Set | 233 |
| Table 14.2-13.2 Raw cumulative incidence of MR 4.0 during post-randomization consolidation phase (ARM 2) by BCR-ABL (IS) ratio at Month 3 - Subset of Full Analysis Set randomized to Arm 2 | 233 |
| Table 14.2-13.2.1 Raw cumulative incidence of MR 4.0 during post-randomization consolidation phase (ARM 2) by BCR-ABL (IS) ratio at Month 3 - Subset of LSC sub-study Full Analysis Set randomized to Arm 2 | 233 |
| Table 14.2-13.3 Raw cumulative incidence of MR 4.0 during re-treatment phase by BCR-ABL (IS) ratio at Month 3 – Subset of Full Analysis Set entering the retreatment phase | 233 |
| Table 14.2-14.1 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase by BCR-ABL (IS) ratio at Month 3 – Full Analysis Set | 234 |
| Table 14.2-14.1.1 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase by BCR-ABL (IS) ratio at Month 3 – LSC sub-study Full Analysis Set | 234 |
| Table 14.2-14.2 Raw cumulative incidence of MR 4.5 during post-randomization consolidation phase (ARM 2) by BCR-ABL (IS) ratio at Month 3 - Subset of Full Analysis Set randomized to Arm 2 | 234 |
| Table 14.2-14.2.1 Raw cumulative incidence of MR 4.5 during post-randomization consolidation phase (ARM 2) by BCR-ABL (IS) ratio at Month 3 - Subset of LSC sub-study Full Analysis Set randomized to Arm 2 | 234 |
| Table 14.2-14.3 Raw cumulative incidence of MR 4.5 during re-treatment phase by BCR-ABL (IS) ratio at Month 3 – Subset of Full Analysis Set entering the retreatment phase | 234 |
| Table 14.2-15.1 Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase by Sokal Risk category– Full Analysis Set2 | |
| Table 14.2-15.2 Raw cumulative incidence of MR4.0 during pre-randomization Induction/Consolidation phase by Sokal Risk category—Full Analysis Set2 | 235 |

| Table 14.2-15.3 Raw cumulative incidence of MR4.5 during pre-randomization Induction/Consolidation phase by Sokal Risk category—Full Analysis Set | .236 |
|---|---|
| Table 14.2-16.1 Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase by time since initial diagnosis of CML–Full Analysis Set | .237 |
| Table 14.2-16.2 Raw cumulative incidence of MR4.0 during pre-randomization Induction/Consolidation phase by time since initial diagnosis of CML – Full Analysis Set | .238 |
| Table 14.2-16.3 Raw cumulative incidence of MR4.5 during pre-randomization Induction/Consolidation phase by time since initial diagnosis of CML – Full Analysis Set | .238 |
| Table 14.2-17.1 Suboptimal response up to 24 months of pre-randomization Induction/Consolidation phase - Full Analysis Set patients who prematurely discontinued the pre-randomization Induction/Consolidation phase | .239 |
| Table 14.2-17.2 Suboptimal response up to 12 months of post-randomization Consolidation phase (ARM 2) - Subset of Full Analysis Set patients who prematurely discontinued the Induction/Consolidation phase randomized to Arm 2 | .240 |
| Table 14.2-18.1 Suboptimal response up to 24 months of pre-randomization Induction/Consolidation phase - Full Analysis Set | .240 |
| Table 14.2-18.2 Suboptimal response up to 12 months of post-randomization Consolidation phase - Subset of Full Analysis Set, randomized to ARM 2 | .240 |
| Table 14.2-19.1 Kinetics of BCR-ABL (IS) ratio during pre-randomization<br>Induction/Consolidation phase – Full Analysis Set | .241 |
| Table 14.2-19.1.1 Kinetics of BCR-ABL (IS) ratio during pre-randomization Induction/Consolidation phase – LSC sub-study Full Analysis Set | .241 |
| Table 14.2-19.2 Kinetics of BCR-ABL (IS) ratio during post-randomization consolidation phase (ARM 2) –Subset of Full Analysis Set randomized to Arm 2 | .242 |
| Table 14.2-19.2.1 Kinetics of BCR-ABL (IS) ratio during post-randomization consolidation phase (ARM 2) –Subset of LSC sub-study Full Analysis Set randomized to Arm 2 | .242 |
| Table 14.2-19.3 Kinetics of BCR-ABL (IS) ratio during TFR phase – Subset of Full Analysis Set entering the TFR phase | .243 |
| Table 14.2-19.4 Kinetics of BCR-ABL (IS) ratio during re-treatment phase – Subset of Full Analysis Set entering the re-treatment phase | |
| Table 14.2-19.5 Kinetics of BCR-ABL (IS) ratio during TFR phase, SDV sensitivity – Subset of Full Analysis Set entering the TFR phase | .246 |
| Table 14.2-19.6 Kinetics of BCR-ABL (IS) ratio during re-treatment phase, SDV sensitivity – Subset of Full Analysis Set entering the re-treatment phase | .246 |
| Table 14.2-20.1 Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase - Full Analysis Set patients not reaching MMR at baseline | 247 |

| Table 14.2-20.2 Raw cumulative incidence of MMR during post-randomization Consolidation phase (ARM 2) - Subset of Full Analysis Set patients not reaching MMR at baseline, randomized to ARM 2 | 247 |
|---|---|
| Table 14.2-21.1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase - Full Analysis Set patients not reaching MR 4.0 at baseline | 247 |
| Table 14.2-21.2 Raw cumulative incidence of MR 4.0 during post-randomization Consolidation phase (ARM 2) - Subset of Full Analysis Set patients not reaching MR 4.0 at baseline, randomized to ARM 2 | 247 |
| Table 14.2-22.1 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase - Full Analysis Set patients not reaching MR 4.5 at baseline | 247 |
| Table 14.2-22.2 Raw cumulative incidence of MR 4.5 during post-randomization Consolidation phase (ARM 2) - Subset of Full Analysis Set patients not reaching MR 4.5 at baseline, randomized to ARM 2 | 248 |
| Table 14.2-22.3 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase - Full Analysis Set patients not reaching MMR at baseline | 248 |
| Table 14.2-22.4 Raw cumulative incidence of MR 4.0 during post-randomization Consolidation phase (ARM 2) - Subset of Full Analysis Set patients not reaching MMR at baseline, randomized to ARM 2 | 248 |
| Table 14.2-22.5 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase - Full Analysis Set patients not reaching MMR at baseline | 248 |
| Table 14.2-22.6 Raw cumulative incidence of MR 4.5 during post-randomization Consolidation phase (ARM 2) - Subset of Full Analysis Set patients not reaching MMR at baseline, randomized to ARM 2 | 248 |
| Table 14.2-23.1 Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase by BCR-ABL(IS) ratio at baseline - Full Analysis Set | 249 |
| Table 14.2-23.1.1 Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase by BCR-ABL (IS) ratio at baseline– LSC substudy Full Analysis Set | |
| Table 14.2-23.2 Raw cumulative incidence of MMR during post-randomization consolidation phase (ARM 2) by BCR-BL(IS) ratio at baseline - Subset of Full Analysis Set, randomized to ARM 2 | 250 |
| Table 14.2-23.2.1 Raw cumulative incidence of MMR during post-randomization consolidation phase (ARM 2) by BCR-BL(IS) ratio at baseline - Subset of LSC sub-study Full Analysis Set , randomized to ARM 2 | 251 |
| Table 14.2-23.3 Raw cumulative incidence of MMR during re-treatment phase by BCR-BL(IS) ratio at baseline – Subset of Full Analysis Set entering the retreatment phase | |
| Table 14.2-24.1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase by BCR-ABL(IS) ratio at baseline - Full Analysis Set | 252 |

| Table 14.2-24.1.1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase by BCR-ABL (IS) ratio at baseline– LSC substudy Full Analysis Set | 52 |
|---|---|
| Table 14.2-24.2 Raw cumulative incidence of MR 4.0 during post-randomization consolidation phase (ARM 2) by BCR-BL(IS) ratio at baseline - Subset of Full Analysis Set, randomized to ARM 2 | 52 |
| Table 14.2-24.2.1 Raw cumulative incidence of MR 4.0 during post-randomization consolidation phase (ARM 2) by BCR-BL(IS) ratio at baseline - Subset of LSC sub-study Full Analysis Set , randomized to ARM 2 | .52 |
| Table 14.2-24.3 Raw cumulative incidence of MR 4.0 during re-treatment phase by BCR-BL(IS) ratio at baseline – Subset of Full Analysis Set entering the retreatment phase | 52 |
| Table 14.2-25.1 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase by BCR-ABL(IS) ratio at baseline - Full Analysis Set | .53 |
| Table 14.2-25.1.1 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase by BCR-ABL (IS) ratio at baseline– LSC substudy Full Analysis Set | .53 |
| Table 14.2-25.2 Raw cumulative incidence of MR 4.5 during post-randomization consolidation phase (ARM 2) by BCR-BL(IS) ratio at baseline - Subset of Full Analysis Set, randomized to ARM 2 | .53 |
| Table 14.2-25.2.1 Raw cumulative incidence of MR 4.5 during post-randomization consolidation phase (ARM 2) by BCR-BL(IS) ratio at baseline - Subset of LSC sub-study Full Analysis Set, randomized to ARM 2 | 53 |
| Table 14.2-25.3 Raw cumulative incidence of MR 4.5 during re-treatment phase by BCR-BL(IS) ratio at baseline – Subset of Full Analysis Set entering the retreatment phase | .53 |
| Table 14.2-26.1 Raw cumulative loss of MMR during TFR phase –Subset of Full Analysis Set entering the TFR phase | 54 |
| Table 14.2-26.2 Raw cumulative loss of MR4.0 during TFR phase –Subset of Full Analysis Set entering the TFR phase —25 | 55 |
| Table 14.2-26.3 Raw cumulative loss of MR4.5 during TFR phase –Subset of Full Analysis Set entering the TFR phase with MR4.5 | 55 |
| Table 14.2-26.4 Raw cumulative loss of MMR during TFR phase, SDV sensitivity – Subset of Full Analysis Set entering the TFR phase | 56 |
| Table 14.2-26.5 Raw cumulative loss of MR4.0 during TFR phase, SDV sensitivity -Subset of Full Analysis Set entering the TFR phase | 56 |
| Table 14.2-26.6 Raw cumulative loss of MR4.5 during TFR phase, SDV sensitivity -Subset of Full Analysis Set entering the TFR phase with MR4.5 | 56 |
| Table 14.2-27.1 Descriptive Statistics for CD34 cells: Total percentage – LSC substudy Full Analysis Set | 57 |
| Table 14.2-28.1 Descriptive Statistics for CD34+/CD38+ cells: Percentage from total CD34+ cells – LSC sub-study Full Analysis Set | 59 |
| Table 14.2-28.2 Descriptive Statistics for number of events sorted in CD34+/CD38+ cells – LSC sub-study Full Analysis Set | 60 |

| Table 14.2-28.3 Ph+ by HIS status, in CD34+/CD38+ cells – LSC sub-study Full Analysis Set |
|---|
| Table 14.2-28.4 Descriptive statistics of Ph+ in CD34+/CD38+ cells- LSC sub-study Full Analysis Set |
| Table 14.2-28.5 BCR-ABL by RT-PCR status, in CD34+/CD38+ cells – LSC substudy Full Analysis Set |
| Table 14.2-29.1 Descriptive Statistics for CD34+/CD38- cells: Percentage from total CD34+ cells – LSC sub-study Full Analysis Set |
| Table 14.2-29.2 Descriptive Statistics for number of events sorted in CD34+/CD38-cells – LSC sub-study Full Analysis Set |
| Table 14.2-29.3 Ph+ by HIS status, in CD34+/CD38- cells – LSC sub-study Full Analysis Set |
| Table 14.2-29.4 Descriptive statistics of Ph+ in CD34+/CD38- cells– LSC sub-study Full Analysis Set |
| Table 14.2-29.5 BCR-ABL by RT-PCR status, in CD34+/CD38- cells – LSC substudy Full Analysis Set |
| Table 14.2-30.1 Descriptive Statistics for Immunophenotypically aberrant CD34+ cells: Percentage from total CD34+ cells –LSC sub-study Full Analysis Set263 |
| Table 14.2-30.2 Descriptive Statistics for number of events sorted in Immunophenotypically aberrant CD34+ cells – LSC sub-study Full Analysis Set |
| Table 14.2-30.3 Ph+ by HIS status, in Immunophenotypically aberrant CD34+ cells - LSC sub-study Full Analysis Set |
| Table 14.2-30.4 Descriptive statistics of Ph+ in Immunophenotypically aberrant CD34+ cells– LSC sub-study Full Analysis Set |
| Table 14.2-30.5 BCR-ABL by RT-PCR status, in Immunophenotypically aberrant CD34+ cells – LSC sub-study Full Analysis Set |
| Table 14.2-31.1 Descriptive Statistics for Immunophenotypically aberrant CD34-cells: Percentage from total CD34+ cells – LSC sub-study Full Analysis Set 264 |
| Table 14.2-31.2 Descriptive Statistics for number of events sorted in Immunophenotypically aberrant CD34- cells- LSC sub-study Full Analysis Set |
| Table 14.2-31.3 Ph+ by HIS status, in Immunophenotypically aberrant CD34- cells – LSC sub-study Full Analysis Set |
| Table 14.2-31.4 Descriptive statistics of Ph+ in Immunophenotypically aberrant CD34- cells- LSC sub-study Full Analysis Set |
| Table 14.2-31.5 BCR-ABL by RT-PCR status, in Immunophenotypically aberrant CD34- cells – LSC sub-study Full Analysis Set |
| Table 14.2-32.1 Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase by duration of prior exposure to Imatinib - Full Analysis Set |
| Table 14.2-32.1.1 Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase by by prior Imatib treatment duration – LSC sub-study Full Analysis Set |

| Table 14.2-32.2 Raw cumulative incidence of MMR during post-randomization consolidation phase (ARM 2) by prior Imatib treatment duration - Subset of Full Analysis Set, randomized to ARM 2 | 266 |
|---|---|
| Table 14.2-32.2.1 Raw cumulative incidence of MMR during post-randomization consolidation phase (ARM 2) by prior Imatib treatment duration - Subset of LSC sub-study Full Analysis Set , randomized to ARM 2 | 267 |
| Table 14.2-32.3 Raw cumulative incidence of MMR during re-treatment phase by prior Imatib treatment duration – Subset of Full Analysis Set entering the retreatment phase | 267 |
| Table 14.2-33.1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase by prior Imatib treatment duration - Full Analysis Set | 268 |
| Table 14.2-33.1.1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase by prior Imatib treatment duration – LSC substudy Full Analysis Set | 268 |
| Table 14.2-33.2 Raw cumulative incidence of MR 4.0 during post-randomization consolidation phase (ARM 2) by prior Imatib treatment duration - Subset of Full Analysis Set, randomized to ARM 2 | 268 |
| Table 14.2-33.2.1 Raw cumulative incidence of MR 4.0 during post-randomization consolidation phase (ARM 2) by prior Imatib treatment duration - Subset of LSC sub-study Full Analysis Set , randomized to ARM 2 | 268 |
| Table 14.2-33.3 Raw cumulative incidence of MR 4.0 during re-treatment phase by prior Imatib treatment duration – Subset of Full Analysis Set entering the retreatment phase | 268 |
| Table 14.2-34.1 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase by prior Imatib treatment duration - Full Analysis Set | 269 |
| Table 14.2-34.1.1 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase by prior Imatib treatment duration – LSC sub- | 269 |
| Table 14.2-34.2 Raw cumulative incidence of MR 4.5 during post-randomization consolidation phase (ARM 2) by prior Imatib treatment duration - Subset of Full Analysis Set, randomized to ARM 2 | 269 |
| Table 14.2-34.2.1 Raw cumulative incidence of MR 4.5 during post-randomization consolidation phase (ARM 2) by prior Imatib treatment duration - Subset of LSC sub-study Full Analysis Set, randomized to ARM 2 | 269 |
| Table 14.2-34.3 Raw cumulative incidence of MR 4.5 during re-treatment phase by prior Imatib treatment duration – Subset of Full Analysis Set entering the retreatment phase | 269 |
| Section 14.3 – Safety data | |
| Table 14.3-1.1 Duration of exposure to study treatment during pre-randomization | 271 |
| Table 14.3-1.1.1 Duration of exposure to study treatment during pre-randomization Induction/Consolidation— LSC sub-study Safety Set | |

| Table 14.3-1.2 Duration of exposure to study treatment during post-randomization Consolidation phase (ARM 2) - Subset of Safety Set randomized to Arm 2272 |
|---|
| Table 14.3-1.2.1 Duration of exposure to study treatment during post-randomization Consolidation phase (ARM 2) - Subset of LSC sub-study Safety Set randomized to Arm 2 |
| Table 14.3-1.1.3 Duration of exposure to study treatment during re-treatment phase – Subset of Safety Set entering the re-treatment phase |
| Table 14.3-1.1.21 Duration of exposure to study treatment during pre-randomization Induction/Consolidation phase, by stable MR4.0 at 24 months and halving time - Safety Set |
| Table 14.3-1.1.22 Duration of exposure to study treatment during pre-randomization Induction/Consolidation phase, by stable MR4.0 by 24 months and halving time - Safety Set |
| Table 14.3-2.1 Relative dose intensity and average daily dose during pre-<br>randomization Induction/Consolidation phase – Safety Set |
| Table 14.3-2.1.1 Relative dose intensity and average daily dose during pre-<br>randomization Induction/Consolidation phase – LSC sub-study Safety Set277 |
| Table 14.3-2.2 Relative dose intensity and average daily dose during post-randomization consolidation phase (ARM 2) – Subset of Safety Set randomized to Arm 2 |
| Table 14.3-2.2.1 Relative dose intensity and average daily dose during post-randomization consolidation phase (ARM 2) – Subset of LSC sub-study Safety Set randomized to Arm 2 |
| Table 14.3-2.3 Relative dose intensity and average daily dose during re-treatment phase – Subset of Safety Set entering the re-treatment phase — 278 |
| Table 14.3-3.1 Dose reduction and interruption during pre-randomization Induction/Consolidation phase - Safety Set |
| Table 14.3-3.1.1 Dose reduction and interruption during pre-randomization Induction/Consolidation phase – LSC sub-study Safety Set |
| Table 14.3-3.2 Dose reduction and interruption during post-randomization consolidation phase (ARM 2) – Subset of Safety Set randomized to Arm 2 280 |
| Table 14.3-3.2.1 Dose reduction and interruption during post-randomization consolidation phase (ARM 2) – Subset of LSC sub-study Safety Set randomized to Arm 2 |
| Table 14.3-3.3 Dose reduction and interruption during re-treatment phase – Subset of Safety Set entering the re-treatment phase |
| Table 14.3-4.1 Concomitant medication by ATC class and preferred term during prerandomization Induction/Consolidation phase Full Analysis Set |
| Table 14.3-4.1.1 Concomitant medication by ATC class and preferred term during pre-randomization Induction/Consolidation phase LSC sub-study Full Analysis Set |
| Table 14.3-4.2 Concomitant medication by ATC class and preferred term during post-randomization consolidation phase (ARM 2)– Subset of Full Analysis Set randomized to Arm 2 |
| Table 14.3-4.2.1 Concomitant medication by ATC class and preferred term during post-randomization consolidation phase (ARM 2)— Subset of LSC sub-study Full Analysis Set randomized to Arm 2 |
|---|
| Table 14.3-4.3 Concomitant medication by ATC class and preferred term during TFR phase – Subset of Full Analysis Set entering the TFR phase |
| Table 14.3-4.4 Concomitant medication by ATC class and preferred term during retreatment phase – Subset of Full Analysis Set entering the re-treatment phase286 |
| Table 14.3-5.1.1 Hematology shift table based on CTCAE grade during Pre-<br>Randomization pre-randomization Induction/Consolidation –Full Analysis<br>Set |
| Table 14.3-5.1.2 Hematology shift table based on CTCAE grade during post-randomization consolidation phase (ARM 2)— Subset of Full Analysis Set randomized to Arm 2 |
| Table 14.3-5.1.3 Hematology shift table based on CTCAE grade during re-treatment phase – Subset of Full Analysis Set entering the re-treatment phase290 |
| Table 14.3-5.1.4 Hematology shift table based on CTCAE grade during whole study period – Full Analysis Set |
| Table 14.3-5.1.5 Hematology shift table based on CTCAE grade during re-treatment phase, SDV sensitivity – Subset of Full Analysis Set entering the retreatment phase |
| Table 14.3-5.1.6 Hematology shift table based on CTCAE grade during whole study period, SDV sensitivity– Full Analysis Set |
| Table 14.3-5.2.1 Biochemistry shift table based on CTCAE grade during post-randomization consolidation phase (ARM 2)— Subset of Full Analysis Set randomized to Arm 2 |
| Table 14.3-5.2.2 Biochemistry shift table based on CTCAE grade during retreatment phase—Subset of Full Analysis Set entering the re-treatment phase294 |
| Table 14.3-5.2.3 Biochemistry shift table based on CTCAE grade during whole study period – Full Analysis Set |
| Table 14.3-5.2.4 Biochemistry shift table based on CTCAE grade during retreatment phase, SDV sensitivity– Subset of Full Analysis Set entering the retreatment phase |
| Table 14.3-5.2.5 Biochemistry shift table based on CTCAE grade during whole study period, SDV sensitivity – Full Analysis Set |
| Table 14.3-6.1.1 Hematology shift table based on normal range for parameters with no defined CTCAE grades during post-randomization consolidation phase (ARM 2)— Subset of Full Analysis Set randomized to Arm 2 |
| Table 14.3-6.1.2 Hematology shift table based on normal range for parameters with no defined CTCAE grades during re-treatment phase – Subset of Full Analysis Set entering the re-treatment phase |
| Table 14.3-6.1.3 Hematology shift table based on normal range for parameters with no defined CTCAE grades during whole study period –Full Analysis Set297 |
| Table 14.3-6.1.4 Hematology shift table based on normal range for parameters with no defined CTCAE grades during re-treatment phase, SDV sensitivity – Subset of Full Analysis Set entering the re-treatment phase |

| Table 14.3-6.1.5 Hematology shift table based on normal range for parameters with no defined CTCAE grades during whole study period, SDV sensitivity –Full Analysis Set | .298 |
|---|---|
| Table 14.3-6.2.1 Biochemistry shift table based on normal range for parameters with no defined CTCAE grades during post-randomization consolidation phase (ARM 2) – Subset of Full Analysis Set randomized to Arm 2 | .299 |
| Table 14.3-6.2.2 Biochemistry shift table based on normal range for parameters with no defined CTCAE grades during re-treatment phase – Subset of Full Analysis Set entering the re-treatment phase | .299 |
| Table 14.3-6.2.3 Biochemistry shift table based on normal range for parameters with no defined CTCAE grades during whole study period –Full Analysis Set | .299 |
| Table 14.3-6.2.4 Biochemistry shift table based on normal range for parameters with no defined CTCAE grades during re-treatment phase, SDV sensitivity – Subset of Full Analysis Set entering the re-treatment phase | .299 |
| Table 14.3-6.2.5 Biochemistry shift table based on normal range for parameters with no defined CTCAE grades during whole study period, SDV sensitivity –Full Analysis Set | .299 |
| Table 14.3-7.1 ECG shift table based on notable values during Pre-randomization Induction Consolidation–Full Analysis Set | .300 |
| Table 14.3-7.2 ECG shift table based on notable values during post-randomization consolidation phase (ARM 2) – Subset of Full Analysis Set randomized to Arm 2 | .301 |
| Table 14.3-7.3 ECG shift table based on notable values during re-treatment phase – Subset of Full Analysis Set entering the re-treatment phase | .302 |
| Table 14.3-7.4 Notable ECG values during pre-randomization Ind/Cons –Full Analysis Set | .303 |
| Table 14.3-7.5 Notable ECG values during post-randomization consolidation phase (ARM 2)— Subset of Full Analysis Set randomized to Arm 2 | .304 |
| Table 14.3-7.6 Notable ECG values during re-treatment phase – Subset of Full Analysis Set entering the re-treatment phase | .305 |
| Table 14.3-7.7 ECG shift table based on notable values during re-treatment phase, SDV sensitivity – Subset of Full Analysis Set entering the re-treatment phase. | .305 |
| Table 14.3-7.8 Notable ECG values during re-treatment phase, SDV sensitivity – Subset of Full Analysis Set entering the re-treatment phase | .305 |
| Table 14.3-8.1 Echocardiography assessment at baseline – Full Analysis Set | .306 |
| Table 14.3-8.2 Echocardiography shift table based on overall interpretation - Full | .307 |
| Table 14.3-8.3 Echocardiography shift table based on overall interpretation, SDV sensitivity - Full Analysis Set | .308 |
| Table 14.3-9.1 Summary statistics of total cholesterol, HDL, LDL, glucose, microalbumin and HbA1c over Induction/Consolidation phase – Full Analysis Set | |
| Table 14.3-9.2.1 Total cholesterol shift table based on specific levels during | 310 |

| Table 14.3-9.2.2 Total cholesterol shift table based on specific levels during TFR phase – Subset of Full Analysis Set entering the TFR phase | 311 |
|---|---|
| Table 14.3-9.2.3 Total cholesterol shift table based on specific levels during Retreatment phase — Subset of Full Analysis Set entering the Re-treatment phase — | |
| Table 14.3-9.2.4 Total cholesterol shift table based on specific levels during TFR phase, SDV sensitivity – Subset of Full Analysis Set entering the TFR phase | |
| Table 14.3-9.2.5 Total cholesterol shift table based on specific levels during Retreatment phase, SDV sensitivity – Subset of Full Analysis Set entering the Re-treatment phase | 312 |
| Table 14.3-10.1.1 Fasting glucose shift table based on specific levels during Induction Consolidation – Full Analysis Set | 313 |
| Table 14.3-10.1.2 Fasting glucose shift table based on specific levels during TFR phase — Subset of Full Analysis Set entering the TFR phase | 314 |
| Table 14.3-10.1.3 Fasting glucose shift table based on specific levels during Retreatment phase — Subset of Full Analysis Set entering the Re-treatment phase — | 314 |
| Table 14.3-10.1.4 Fasting glucose shift table based on specific levels during TFR phase, SDV sensitivity — Subset of Full Analysis Set entering the TFR phase. | 314 |
| Table 14.3-10.1.5 Fasting glucose shift table based on specific levels during Retreatment phase, SDV sensitivity — Subset of Full Analysis Set entering the Re-treatment phase | 315 |
| Table 14.3-11.1 Vital Signs during Induction Consolidation – Full Analysis Set | 316 |
| Table 14.3-11.2 Vital Signs during TFR phase – Subset of Full Analysis Set entering the TFR phase | 319 |
| Table 14.3-11.3 Vital Signs during Re-treatment phase — Subset of Full Analysis Set entering the Re-treatment phase — | 319 |
| Table 14.3-11.4 Vital Signs during TFR phase, SDV sensitivity – Subset of Full Analysis Set entering the TFR phase. | 320 |
| Table 14.3-11.5 Vital Signs during Re-treatment phase, SDV sensitivity – Subset of Full Analysis Set entering the Re-treatment phase | 320 |
| Table 14.3-12.1 Survival follow-up – Full Analysis Set. | 321 |
| Table 14.3-12.2 Survival follow-up, SDV sensitivity – Full Analysis Set | 322 |
| Table 14.3-13.1 Safety follow-up – Full analysis Set | 323 |
| Table 14.3-13.2 Safety follow-up, SDV sensitivity – Full analysis Set | 323 |
| Section 14.3.1 – Displays of adverse events | 324 |
| Figure 14.3.1-1.1 Kaplan-Meier analysis of time-to-first CVEs during the pre-<br>randomization Induction/Consolidation phase – Full Analysis Set | 324 |
| Figure 14.3.1-1.2 Kaplan-Meier analysis of time-to-first CVEs during the post-randomization consolidation phase (ARM 2) – Subset of Full Analysis Set randomized to Arm 2 | 325 |
| Figure 14.3.1-1.3 Kaplan-Meier analysis of time-to-first CVEs during the the TFR phase – Subset of Full Analysis Set entering the TFR phase | 326 |

| Figure | 14.3.1-1.4 Kaplan-Meier analysis of time-to-first CVEs during the retreatment phase – Subset of Full Analysis Set entering the re-treatment phase | .326 |
|---|---|---|
| Figure | 14.3.1-2.1 Number of sorted events by HIS CD34+/CD38+ cells | .327 |
| Figure | 14.3.1-2.2 Number of sorted events by PCR CD34+/CD38+ cells | .328 |
| Figure | 14.3.1-3.1 Number of sorted events by HIS CD34+/CD38- cells | .328 |
| Figure | 14.3.1-3.2 Number of sorted events by PCR CD34+/CD38- cells | .328 |
| Figure | 14.3.1-4.1 Number of sorted events by HIS Immunophenotypically aberrant CD34+ cells | .328 |
| Figure | 14.3.1-4.2 Number of sorted events by PCR Immunophenotypically aberrant CD34+ cells | .328 |
| Figure | 14.3.1-5.1 Number of sorted events by HIS Immunophenotypically aberrant CD34- cells | .328 |
| Figure | 14.3.1-5.2 Number of sorted events by PCR Immunophenotypically aberrant CD34- cells | .328 |
| Figure | 14.3.1-6.1 Number of HIS+ subjects CD34+/CD38+ cells – LSC substudy Full Analysis Set | .329 |
| Figure | 14.3.1-6.2 Number of PCR subjects CD34+/CD38+ cells – LSC substudy Full Analysis Set | .330 |
| _ | 14.3.1-7.1 Number of HIS+ subjects CD34+/CD38- cells – LSC substudy Full Analysis Set | .330 |
| Figure | 14.3.1-7.2 Number of PCR subjects CD34+/CD38- cells – LSC substudy Full Analysis Set | .330 |
| Figure | 14.3.1-8.1 Number of HIS+ subjects Immunophenotypically aberrant CD34+ cells – LSC substudy Full Analysis Set | .330 |
| Figure | 14.3.1-8.2 Number of PCR subjects Immunophenotypically aberrant CD34+ cells – LSC substudy Full Analysis Set | .330 |
| Figure | 14.3.1-9.1 Number of HIS+ subjects Immunophenotypically aberrant CD34-cells – LSC substudy Full Analysis Set | .330 |
| Figure | 14.3.1-9.2 Number of PCR subjects Immunophenotypically aberrant CD34-cells – LSC substudy FAS | .330 |
| Figure | 14.3.1-10 Number of patients with detectable LSC – LSC substudy Full Analysis Set | .331 |
| Table 1 | 14.3.1-1.1 Overall summary of treatment-emergent adverse events occurring during pre-randomization Induction/consolidation phase – Full Analysis Set | .332 |
| Table 1 | 14.3.1-1.2 Overall summary of treatment-emergent adverse events occurring during post-randomization consolidation phase (ARM 2) – Subset of Full Analysis Set randomized to Arm 2 | .334 |
| Table 1 | 14.3.1-1.3 Overall summary of treatment-emergent adverse events occurring during re-treatment phase — Subset of Full Analysis Set entering the retreatment phase | .336 |
| Table 1 | 14.3.1-1.4 Overall summary of adverse events occurring during TFR phase – Subset of Full Analysis Set entering the TFR phase | .337 |

| Table 14.3.1-2.1 Overall summary of frequent [1] treatment-emergent adverse events occurring during pre-randomization Induction/consolidation phase – Full Analysis Set | .338 |
|---|---|
| Table 14.3.1-2.2 Overall summary of frequent [1] treatment-emergent adverse events occurring during post-randomization consolidation phase (ARM 2) – Subset of Full Analysis Set randomized to Arm 2 | |
| Table 14.3.1-2.3 Overall summary of frequent [1] treatment-emergent adverse events occurring during re-treatment phase — Subset of Full Analysis Set entering the re-treatment phase | .338 |
| Table 14.3.1-2.4 Overall summary of frequent [1] adverse events occurring during TFR phase – Subset of Full Analysis Set entering the TFR phase | .339 |
| Table 14.3.1-3.1.1 Treatment Emergent adverse events incidence, regardless of study drug relationship, occurring during pre-randomization Induction/consolidation phase by system organ class and preferred term - overall and maximum grade 3/4 – Full Analysis Set | .340 |
| Table 14.3.1-3.1.2 Treatment Emergent adverse events occurence, regardless of study drug relationship, occurring during pre-randomization Induction/consolidation phase by system organ class and preferred term - overall and maximum grade 3/4 – Full Analysis Set | .341 |
| Table 14.3.1-3.2.1 Treatment Emergent adverse events incidence, regardless of study drug relationship, occurring during post-randomization consolidation phase (ARM 2) by system organ class and preferred term - overall and maximum grade 3/4 – Subset of Full Analysis Set randomized to Arm 2 | |
| Table 14.3.1-3.2.2 Treatment Emergent adverse events occurence, regardless of study drug relationship, occurring during post-randomization consolidation phase (ARM 2) by system organ class and preferred term - overall and maximum grade 3/4 – Subset of Full Analysis Set randomized to Arm 2 | .343 |
| Table 14.3.1-3.3.1 Treatment-emergent adverse events incidence, regardless of study drug relationship, by system organ class and preferred term during retreatment phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the re-treatment phase | .344 |
| Table 14.3.1-3.3.2 Treatment-emergent adverse events occurrence, regardless of study drug relationship, by system organ class and preferred term during retreatment phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the re-treatment phase | .345 |
| Table 14.3.1-3.4.1 Adverse events incidence, regardless of study drug relationship, by system organ class and preferred term during TFR phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the TFR phase | .345 |
| Table 14.3.1-3.4.2 Adverse events occurrence, regardless of study drug relationship, by system organ class and preferred term during TFR phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the TFR phase | .345 |
| Table 14.3.1-3.5.1 Frequent [1] Treatment Emergent adverse events incidence, regardless of study drug relationship occurring during pre-randomization Induction/consolidation phase by system organ class and preferred term | 246 |
| overall and maximum grade 3/4 – Full Analysis Set | .346 |

| Table 14.3.1-3.5.2 Frequent [1] Treatment Emergent adverse events incidence, regardless of study drug relationship occurring during post-randomization consolidation phase (ARM 2) by system organ class and preferred termoverall and maximum grade 3/4 – Subset of Full Analysis Set randomized to Arm 2 | to<br>346 |
|---|---|
| Table 14.3.1-3.5.3 Frequent [1] Treatment Emergent adverse events incidence, regardless of study drug relationship occurring during re-treatment phase by system organ class and preferred term- overall and maximum grade 3/4 – Subset of Full Analysis Set entering the re-treatment phase | |
| Table 14.3.1-3.5.4 Frequent [1] adverse events incidence, regardless of study drug relationship occurring during TFR phase by system organ class and preferre term - overall and maximum grade 3/4 – Subset of Full Analysis Set entering the TFR phase | |
| Table 14.3.1-4.1.1 Serious treatment-emergent adverse events incidence, regardless of study drug relationship, by system organ class and preferred term during pre-randomization Induction/consolidation phase – overall and maximum grade 3/4 –Full Analysis Set | 348 |
| Table 14.3.1-4.1.2 Serious treatment-emergent adverse events occurence, regardles of study drug relationship, by system organ class and preferred term during pre-randomization Induction/consolidation phase – overall and maximum grade 3/4 –Full Analysis Set | 348 |
| Table 14.3.1-4.2.1 Serious treatment-emergent adverse events incidence, regardless of study drug relationship, by system organ class and preferred term during post-randomization consolidation phase (ARM 2) – overall and maximum grade 3/4 – Subset of Full Analysis Set randomized to Arm 2 | 349 |
| Table 14.3.1-4.2.2 Serious treatment-emergent adverse events occurrence, regardle of study drug relationship, by system organ class and preferred term during post-randomization consolidation phase (ARM 2) – overall and maximum grade 3/4 – Subset of Full Analysis Set randomized to Arm 2 | ss<br>349 |
| Table 14.3.1-4.3.1 Serious treatment-emergent adverse events incidence, regardless of study drug relationship, by system organ class and preferred term during re-treatment phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the re-treatment phase | |
| Table 14.3.1-4.3.2 Serious treatment-emergent adverse events occurrence, regardle of study drug relationship, by system organ class and preferred term during re-treatment phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the re-treatment phase | |
| Table 14.3.1-4.4.1 Serious adverse events incidence, regardless of study drug relationship, by system organ class and preferred term during TFR phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the TFR phase | 350 |
| Table 14.3.1-4.4.2 Serious adverse events occurence, regardless of study drug relationship, by system organ class and preferred term during TFR phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the TFR phase | |
| Table 14.3.1-4.5.1 Frequent [1] Serious Treatment Emergent adverse events incidence, regardless of study drug relationship occurring during pre- | |

| randomization Induction/consolidation phase by system organ class and preferred term - overall and maximum grade 3/4 – Full Analysis Set | 351 |
|---|---|
| Table 14.3.1-4.5.2 Frequent [1] Serious Treatment Emergent adverse events incidence, regardless of study drug relationship occurring during post-randomization consolidation phase (ARM 2) by system organ class and preferred term - overall and maximum grade 3/4 — Subset of Full Analysis Set randomized to Arm 2 | 351 |
| Table 14.3.1-4.5.3 Frequent [1] Serious Treatment Emergent adverse events incidence, regardless of study drug relationship occurring during re-treatment phase by system organ class and preferred term - overall and maximum grade 3/4 – Subset of Full Analysis Set entering the re-treatment phase | 351 |
| Table 14.3.1-4.5.4 Frequent [1] Serious adverse events incidence, regardless of study drug relationship occurring during TFR phase by system organ class and preferred term - overall and maximum grade 3/4 — Subset of Full Analysis Set entering the TFR phase | 351 |
| Table 14.3.1-4.6.1 Serious treatment-emergent adverse events incidence, suspected to be study drug related, by system organ class and preferred term during prerandomization Induction/consolidation phase — overall and maximum grade 3/4—Full Analysis Set | 352 |
| Table 14.3.1-4.6.2 Serious treatment-emergent adverse events occurence, suspected to be study drug related, by system organ class and preferred term during prerandomization Induction/consolidation phase – overall and maximum grade 3/4 –Full Analysis Set | 352 |
| Table 14.3.1-4.7.1 Serious treatment-emergent adverse events incidence, suspected to be study drug related, by system organ class and preferred term during post-randomization consolidation phase (ARM 2) – overall and maximum grade 3/4 – Subset of Full Analysis Set randomized to Arm 2 | 353 |
| Table 14.3.1-4.7.2 Serious treatment-emergent adverse events occurrence, suspected to be study drug related, by system organ class and preferred term during post-randomization consolidation phase (ARM 2) – overall and maximum grade 3/4 – Subset of Full Analysis Set randomized to Arm 2 | 353 |
| Table 14.3.1-4.8.1 Serious treatment-emergent adverse events incidence, suspected to be study drug related, by system organ class and preferred term during retreatment phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the re-treatment phase | 353 |
| Table 14.3.1-4.8.2 Serious treatment-emergent adverse events occurrence, suspected to be study drug related, by system organ class and preferred term during retreatment phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the re-treatment phase | 353 |
| Table 14.3.1-4.9.1 Serious adverse events incidence, suspected to be study drug related, by system organ class and preferred term during TFR phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the TFR phase | 353 |
| Table 14.3.1-4.9.2 Serious adverse events occurrence, suspected to be study drug related, by system organ class and preferred term during TFR phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the TFR | 354 |

| Table 14.3.1-5.1.1 Treatment-emergent adverse events incidence leading to study drug discontinuation by system organ class and preferred term during prerandomization Induction/Consolidation phase – overall and maximum grade 3/4 –Full Analysis Set | 354 |
|---|---|
| Table 14.3.1-5.1.2 Treatment-emergent adverse events occurence leading to study drug discontinuation by system organ class and preferred term during prerandomization Induction/Consolidation phase – overall and maximum grade 3/4 –Full Analysis Set | 355 |
| Table 14.3.1-5.2.1 Treatment-emergent adverse events incidence leading to study drug discontinuation by system organ class and preferred term during post-randomization phase (ARM 2) – overall and maximum grade 3/4 – Subset of Full Analysis Set randomized to Arm 2 | 355 |
| Table 14.3.1-5.2.2 Treatment-emergent adverse events occurrence leading to study drug discontinuation by system organ class and preferred term during post-randomization phase (ARM 2)— overall and maximum grade 3/4 — Subset of Full Analysis Set randomized to Arm 2 | 355 |
| Table 14.3.1-5.3.1 Treatment-emergent adverse events incidence leading to study drug discontinuation by system organ class and preferred term during retreatment phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the re-treatment phase | 356 |
| Table 14.3.1-5.3.2 Treatment-emergent adverse events occurrence leading to study drug discontinuation by system organ class and preferred term during retreatment phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the re-treatment phase | 356 |
| Table 14.3.1-6.1.1 Treatment-emergent adverse events incidence requiring dosage adjustment or temporarily interruption by system organ class and preferred term during pre-randomization Induction/ consolidation phase — overall and maximum grade 3/4 —Full Analysis Set | 356 |
| Table 14.3.1-6.1.2 Treatment-emergent adverse events occurrence requiring dosage adjustment or temporarily interruption by system organ class and preferred term during pre-randomization Induction/consolidation phase – overall and maximum grade 3/4 –Full Analysis Set | 357 |
| Table 14.3.1-6.2.1 Treatment-emergent adverse events incidence requiring dosage adjustment or temporarily interruption by system organ class and preferred term during post-randomization consolidation phase (ARM 2) – overall and maximum grade 3/4 – Subset of Full Analysis Set randomized to Arm 2 | 357 |
| Table 14.3.1-6.2.2 Treatment-emergent adverse events occurrence requiring dosage adjustment or temporarily interruption by system organ class and preferred term during post-randomization consolidation phase (ARM 2) – overall and maximum grade 3/4 – Subset of Full Analysis Set randomized to Arm 2 | 357 |
| Table 14.3.1-6.3.1 Treatment-emergent adverse events incidence requiring dosage adjustment or temporarily interruption by system organ class and preferred term during re-treatment phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the re-treatment phase | |
| Table 14.3.1-6.3.2 Treatment-emergent adverse events occurrence requiring dosage adjustment or temporarily interruption by system organ class and preferred | |

| term during re-treatment phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the re-treatment phase | |
|---|---|
| Table 14.3.1-6.4.1 Treatment-emergent adverse events of interest incidence, regardless of study drug relationship, by specific group and preferred term during Pre-randomization Induction/consolidation phase –by treatment arm overall and maximum grade 3/4 – Full Analysis Set | |
| Table 14.3.1-6.4.2 Treatment-emergent adverse events of interest occurrence, regardless of study drug relationship, by specific group and preferred term during Pre-randomization Induction/consolidation phase – by treatment arm overall and maximum grade 3/4 –Full Analysis Set | |
| Table 14.3.1-6.5.1 Treatment-emergent adverse events of interest incidence by specific group and preferred term during post-randomization consolidation phase (ARM 2) – overall and maximum grade 3/4 – Subset of Full Analysis Set randomized to Arm 2 | |
| Table 14.3.1-6.5.2 Treatment-emergent adverse events of interest occurrence, by specific group and preferred term during post-randomization consolidation phase (ARM 2) – overall and maximum grade 3/4 – Subset of Full Analysis Set randomized to Arm 2 | |
| Table 14.3.1-6.6.1 Treatment-emergent adverse events of interest incidence by specific group and preferred term during re-treatment phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the re-treatment phase | |
| Table 14.3.1-6.6.2 Treatment-emergent adverse events of interest occurrence by specific group and preferred term during re-treatment phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the re-treatment phase | |
| Table 14.3.1-6.7.1 Adverse events of interest incidence by specific group and preferred term during TFR phase – overall and maximum grade 3/4 – Subse of Full Analysis Set entering the TFR phase | |
| Table 14.3.1-6.7.2 Adverse events of interest occurrence by specific group and preferred term during TFR phase – overall and maximum grade 3/4 – Subse of Full Analysis Set entering the TFR phase | |
| Table 14.3.1-7.1.1 Treatment Emergent adverse events of interest incidence, regardless of study drug relationship, by specific group and preferred term and by cardiovascular risk factors during Pre-randomization Induction/consolidation phase – by treatment arm, overall and maximum grade 3/4 – Full Analysis Set | 365 |
| Table 14.3.1-7.1.2 Treatment Emergent adverse events of interest occurrence, regardless of study drug relationship, by specific group and preferred term and by cardiovascular risk factors during Pre-randomization Induction/consolidation phase – by treatment arm, overall and maximum grade 3/4 –Full Analysis Set | 366 |
| Table 14.3.1-7.2.1 Treatment-emergent adverse events of interest incidence, regardless of study drug relationship, during post-randomization consolidation phase (ARM 2), by specific group and preferred term, and by cardiovascular risk factor—overall and maximum grade 3 or 4 — Subset of Full Analysis Set randomized to Arm 2 | 367 |

| Table 14.3.1-7.2.2 Treatment-emergent adverse events of interest occurrence, regardless of study drug relationship, during post-randomization consolidation phase (ARM 2), by specific group and preferred term, and by cardiovascular risk factor – overall and maximum grade 3 or 4 – Subset of Full Analysis Set randomized to Arm 2 | .368 |
|---|---|
| Table 14.3.1-7.3.1 Treatment-emergent adverse events of interest incidence, regardless of study drug relationship, during re-treatment phase, by specific group and preferred term, and by cardiovascular risk factor – Subset of Full | .369 |
| Table 14.3.1-7.3.2 Treatment-emergent adverse events of interest occurrence, regardless of study drug relationship, during re-treatment phase, by specific group and preferred term, and by cardiovascular risk factor – Subset of Full Analysis Set entering the re-treatment phase. | .370 |
| Table 14.3.1-7.4.1 Adverse events of interest incidence, regardless of study drug relationship, during TFR phase, by specific group and preferred term, and by cardiovascular risk factor – Subset of Full Analysis Set entering the TFR phase | .371 |
| Table 14.3.1-7.4.2 Adverse events of interest occurrence, regardless of study drug relationship, during TFR phase, by specific group and preferred term, and by cardiovascular risk factor – Subset of Full Analysis Set entering the TFR phase | .371 |
| Table 14.3.1-7.5.1 Treatment-emergent adverse events of interest incidence, regardless of study drug relationship, during pre-randomization Induction/consolidation phase, by specific group and preferred term and by 4 cardiovascular risk factors – overall and maximum grade 3/4 –Full Analysis Set | .372 |
| Table 14.3.1-7.5.2 Treatment-emergent adverse events of interest occurence, regardless of study drug relationship, during pre-randomization Induction/consolidation phase, by specific group and preferred term and by 4 cardiovascular risk factors – overall and maximum grade 3/4 –Full Analysis | .372 |
| Table 14.3.1-7.6.1 Treatment-emergent adverse events of interest incidence, regardless of study drug relationship, during post-randomization consolidation phase (ARM 2), by specific group and preferred term, and by 4 categories of cardiovascular risk factors— overall and maximum grade 3 or 4—Subset of Full Analysis Set randomized to Arm 2 | |
| Table 14.3.1-7.6.2 Treatment-emergent adverse events of interest occurrence, regardless of study drug relationship, during post-randomization consolidation phase (ARM 2), by specific group and preferred term, and by 4 categories of cardiovascular risk factors – overall and maximum grade 3 or 4 – Subset of Full Analysis Set randomized to Arm 2 | .372 |
| Table 14.3.1-7.7.1 Treatment-emergent adverse events of interest incidence, regardless of study drug relationship, during re-treatment phase, by specific group and preferred term, and by 4 categories of cardiovascular risk factors – Subset of Full Analysis Set entering the re-treatment phase | .373 |
| Table 14.3.1-7.7.2 Treatment-emergent adverse events of interest occurrence, regardless of study drug relationship, during re-treatment phase, by specific | |

| group and preferred term, and by 4 categories of cardiovascular risk factors—Subset of Full Analysis Set entering the re-treatment phase | .373 |
|---|---|
| Table 14.3.1-7.8.1 Adverse events of interest incidence, regardless of study drug relationship, during TFR phase, by specific group and preferred term, and by 4 categories of cardiovascular risk factors – Subset of Full Analysis Set entering the TFR phase | .374 |
| Table 14.3.1-7.8.2 Adverse events of interest occurrence, regardless of study drug relationship, during TFR phase, by specific group and preferred term, and by 4 categories of cardiovascular risk factors—Subset of Full Analysis Set entering the TFR phase | .374 |
| Table 14.3.1-9.1 On treatment deaths, by system organ class and preferred term during pre-randomization Induction/Consolidation phase - Safety Set | .375 |
| Table 14.3.1-9.2 On treatment deaths, by system organ class and preferred term during post-randomization consolidation phase (ARM 2) – Subset of Safety Set randomized to Arm 2 | .376 |
| Table 14.3.1-9.3 On treatment deaths, by system organ class and preferred term during re-treatment phase – Subset of Safety Set entering the re-treatment phase | .376 |
| Table 14.3.1-10.1.1 Cardiac and vascular adverse events of interest, incidence, by treatment arm during the pre-randomization induction/consolidation phase - Full Analysis Set | .377 |
| Table 14.3.1-10.1.2 Cardiac and vascular adverse events of interest, occurence, by treatment arm during the pre-randomization induction/consolidation phase - Full Analysis Set | .379 |
| Table 14.3.1-10.2.1 Cardiac and vascular adverse events of interest incidence, during the post-randomization consolidation phase (ARM 2) - Subset of Full Analysis Set randomized to Arm 2 | .380 |
| Table 14.3.1-10.2.2 Cardiac and vascular adverse events of interest occurrence, during the post-randomization consolidation phase (ARM 2) - Subset of Full Analysis Set randomized to Arm 2 | .381 |
| Table 14.3.1-10.3.1 Cardiac and vascular adverse events of interest, incidence, by treatment arm during the re-treatment phase — Subset of Full Analysis Set entered re-treatment phase | .381 |
| Table 14.3.1-10.3.2 Cardiac and vascular adverse events of interest, occurence, by treatment arm during the re-treatment phase - Subset of Full Analysis Set entered re-treatment phase | .382 |
| Table 14.3.1-10.4.1 Cardiac and vascular adverse events of interest, incidence, by treatment arm during the TFR phase – Subset of Full Analysis Set entered TFR phase | .383 |
| Table 14.3.1-10.4.2 Cardiac and vascular adverse events of interest, occurence, by treatment arm during the TFR phase - Subset of Full Analysis Set entered TFR phase | |
| Table 14.3.1-10.5 Relationship between cardiac and vascular adverse events of interest with total cholesterol values - Full Analysis Set | |
| Table 14.3.1-10.6 Relationship between cardiac and vascular adverse events of interest with glycemic values - Full Analysis Set | .385 |

| Table 14.3.1-11.1.1 Kaplan-Meier estimate of time-to-first CVEs during the pre-<br>randomization induction/consolidation phase – Full analysis set | .386 |
|---|---|
| Table 14.3.1-11.1.2 Kaplan-Meier estimate of time-to-first CVEs during the post-randomization consolidation phase (ARM 2)— Subset of Full Analysis Set patients randomized on Arm 2 | .389 |
| Table 14.3.1-11.2 Kaplan-Meier estimate of time-to-first CVEs during the retreatment phase – Subset of Full Analysis Set entering the re-treatment phase | .390 |
| Table 14.3.1-12.1 Medical history by system organ class and preferred term- Full Analysis Set | .391 |
| Table 14.3.1-13.1 Prior exposure to imatinib before screening, MMR, age, and Sokal by LSC detection category - LSC sub-study Full Analysis Set | .392 |
| Table 14.3.1-13.2.1 Percentage from total CD34+ cells, CD34+/CD38+ cells - Subgroup of LSC sub-study Full Analysis Set, LSC detected | .393 |
| Table 14.3.1-13.2.2 Percentage from total CD34+ cells, CD34+/CD38- cells - Subgroup of LSC sub-study Full Analysis Set, LSC detected | .394 |
| Table 14.3.1-13.2.3 Percentage from total CD34+ cells, Immunophenotypically aberrant CD34+ cells - Subgroup of LSC sub-study Full Analysis Set, LSC detected | .394 |
| Table 14.3.1-13.2.4 Percentage from total CD34+ cells, Immunophenotypically aberrant CD34 negative cells - Subgroup of LSC sub-study Full Analysis Set, LSC detected | .395 |
| Table 14.3.1-13.3.1 Percentage of Ph+ cells, CD34+/CD38- cells - Subgroup of LSC sub-study Full Analysis Set, LSC detected | .395 |
| Table 14.3.1-13.3.2 Percentage of Ph+ cells, CD34+/CD38- cells - Subgroup of LSC sub-study Full Analysis Set, LSC detected | .395 |
| Table 14.3.1-13.3.3 Percentage of Ph+ cells, Immunophenotypically aberrant CD34+ cells - Subgroup of LSC sub-study Full Analysis Set, LSC detected | .395 |
| Table 14.3.1-13.3.4 Percentage of Ph+ cells, Immunophenotypically aberrant CD34 negative cells - Subgroup of LSC sub-study Full Analysis Set, LSC detected | .395 |
| Table 14.3.1-13.4 Total Percentage of CD34+ cells- Subgroup of LSC sub-study Full Analysis Set, LSC detected | |
| Table 14.3.1-13.5 LSC detection - LSC sub-study Full Analysis Set | .396 |
| Section 14.3.2 – Listings of deaths, other serious and significant adverse events | .397 |
| Listing 14.3.2-1.1 Listing of deaths – Full Analysis Set | .397 |
| Listing 14.3.2-1.2 Listing of deaths SDV sensitivity – Full Analysis Set | .397 |
| Listing 14.3.2-2.1 Listing of adverse events of special interest – Full Analysis Set | .398 |
| Listing 14.3.2-2.2 Listing of adverse events leading to study drug discontinuation – Full Analysis Set | .398 |
| Listing 14.3.2-2.3 Listing of adverse events leading to study drug discontinuation during re-treatment phase – Subset of Full Analysis Set entering the retreatment period | .399 |
| Section 14.3.3 – Narratives of deaths, other serious and significant adverse events (non statistics and programming deliverables) | |
| Section 14.3.4 – Abnormal laboratory value listings | |

| Listing 14.3.4-1.1 Listing of abnormal hematology laboratory value – Full Analysis Set |
|---|
| Listing 14.3.4-2.1 Listing of abnormal biochemistry laboratory value – Full Analysis Set |
| Section 16 – Appendices 40 |
| Section 16.1 – Study information |
| Section 16.1.6 – Listing of patients receiving test drug(s)/investigational product(s) from specific batches where more than one batch was used |
| Section 16.1.7 – Randomization scheme and codes (subject identification and treatment assigned) |
| Listing 16.1.7-1.1 Randomization schemes - Randomized patients40 |
| Section 16.1.9 – Documentation of statistical methods40 |
| Listing 16.1.9.1 Raw Statistical output from Demographic and characteristics at baseline– Full Analysis Set |
| Listing 16.1.9.1.1 Raw Statistical output from Demographic and characteristics at baseline– LSC sub-study Full Analysis Set |
| Listing 16.1.9.2 Raw Statistical output from History of prior Imatinib therapy – Full Analysis Set |
| Listing 16.1.9.2.1 Raw Statistical output from History of prior Imatinib therapy – LSC sub-study Full Analysis Set40 |
| Listing 16.1.9.3 Raw Statistical output from Cardiovascular risk factors at baseline - Full Analysis Set40 |
| Listing 16.1.9.4.1 Raw Statistical output from Molecular response MR4.0 at 12 months of TFR–Subset of Full Analysis Set entering the TFR phase40 |
| Listing 16.1.9.4.2 Raw Statistical output from Molecular response MR4.0 at 12 months of TFR-Subset of Per Protocol Analysis Set entering the TFR phase 40 |
| Listing 16.1.9.5.1 Raw Statistical output from Kaplan-Meier analysis of treatment-free survival during the TFR phase – Subset of Full Analysis Set entering the TFR phase |
| Listing 16.1.9.5.2 Raw Statistical output from Kaplan-Meier analysis of treatment-free survival during the TFR phase – Subset of Per Protocol Analysis Set entering the TFR phase |
| Listing 16.1.9.5.3 Raw Statistical output from Kaplan-Meier analysis of overall survival from Randomization–Randomized Set |
| Listing 16.1.9.5.4 Raw Statistical output from Kaplan-Meier analysis of progression-free survival during the TFR phase – Subset of Full Analysis Set entering the TFR phase |
| Listing 16.1.9.6.1 Raw Statistical output from Kaplan-Meier estimate of time-to-first CVEs during the pre-randomization induction/consolidation phase – Full analysis set |
| Listing 16.1.9.6.2 Raw Statistical output from Kaplan-Meier estimate of time-to-<br>first CVEs during the post-randomization consolidation phase (ARM 2)—<br>Subset of Full Analysis Set patients randomized on Arm 2 |

| Listing 16.1.9.6.3 Raw Statistical output from Kaplan-Meier estimate of time-to-first CVEs during the re-treatment phase – Subset of Full Analysis Set entering the re-treatment phase | 407 |
|---|---|
| Section 16.2 – Patient data listings | |
| Listing 16.2-1.1 Enrolled patients | |
| Section 16.2.1 – Discontinued subjects | |
| Listing 16.2.1-1.1 Treatment and study completion - Safety Set | |
| Listing 16.2.1-1.2 Study discontinuation – Full Analysis Set | |
| Listing 16.2.1-1.3 Screen failures (All subjects enrolled) | |
| Section 16.2.2 – Protocol deviations | |
| Listing 16.2.2-1.1 Protocol deviations – Enrolled patients | |
| Section 16.2.3 – Patients excluded from the efficacy analysis | |
| Listing 16.2.3-1.1 Analysis set – All patients | |
| Section 16.2.4 – Demographics and data at screening | 415 |
| Listing 16.2.4-1.1 Demographic data – Full Analysis Set | 415 |
| Listing 16.2.4-2.1 Family history – Full Analysis Set | 415 |
| Listing 16.2.4-2.2 Disease history– Full Analysis Set | 416 |
| Listing 16.2.4-3.1 Disease history I– Full Analysis Set | 417 |
| Listing 16.2.4-3.2 Disease history II– Full Analysis Set | 418 |
| $Listing \ 16.2.4-3.3 Medical \ history/current \ medical \ condition-Full \ Analysis \ Set \dots$ | 418 |
| Listing 16.2.4.4 Cardiovascular risk factors at baseline for patients with not evaluable CV risk factor, Full Analysis Set | 419 |
| Section 16.2.5 – Compliance and/or drug concentration data if available (including Bioanalytical Data Report) | 420 |
| Listing 16.2.5-1.1 Dosage administration records – Full Analysis Set | 420 |
| Section 16.2.6 – Individual efficacy response data | 420 |
| Listing 16.2.6-1.1 BCR-ABL(IS) ratio and molecular responses during Induction/Consolidation and post-randomization consolidation phase (ARM 2) – Full Analysis Set | 420 |
| Listing 16.2.6-1.2 BCR-ABL(IS) ratio and molecular responses during TFR phase – Subset of Full Analysis Set entering the TFR phase | |
| Listing 16.2.6-1.3 BCR-ABL(IS) ratio and molecular responses during re-treatment phase – Subset of Full Analysis Set entering the re-treatment phase | 421 |
| Listing 16.2.6-2.1 Criteria of successful TFR – Subset of Full Analysis Set entering the TFR phase | 422 |
| Listing 16.2.6-3.1 Assessment of progression-free survival during the TFR phase – Subset of Full Analysis Set entering the TFR phase | 423 |
| Listing 16.2.6-3.2 Assessment of treatment-free survival during the TFR phase – Subset of Full Analysis Set entering the TFR phase | |
| Listing 16.2.6-3.3 Assessment of overall survival From Randomization – | 425 |

| Listing 16.2.6-3.4 Assessment of relapse and treatment status during the TFR phase -Subset of Full Analysis Set entering the TFR phase and relapsed | 426 |
|---|---|
| Listing 16.2.6-4.1 WBC and molecular response in patients with WBC increase (CTCAE grade>G1) – Full Analysis Set | 427 |
| Listing 16.2.6-5.1 Individual Efficacy data, Molecular response – Full Analysis Set. | 428 |
| Listing 16.2.6-5.2 Individual Efficacy data, Bone-marrow I – Full Analysis Set | |
| Listing 16.2.6-5.3 Individual Efficacy data, Bone -marrow II – Full Analysis Set | |
| Listing 16.2.6-6.1.1 Total percentage of CD34+ cells – LSC sub-study Full Analysis Set | 431 |
| Listing 16.2.6-6.2.1 Percentage of cells from total CD34 positive— LSC sub-study Full Analysis Set | 432 |
| Listing 16.2.6-6.3.1 Number of events sorted– LSC sub-study Full Analysis Set | 433 |
| Listing 16.2.6-6.4.1 Ph+ by HIS- LSC sub-study Full Analysis Set | 434 |
| Listing 16.2.6-6.5.1 BCR-ABL by RT-PCR-LSC sub-study Full Analysis Set | 435 |
| Section 16.2.7 – Adverse event listings | 436 |
| Listing 16.2.7-1.1 All adverse events – Full Analysis Set | 436 |
| Listing 16.2.7-2.1 Serious adverse events Full Analysis Set | 437 |
| Listing 16.2.7-2.2 Adverse events leading to study drug discontinuation – Full Analysis Set | 438 |
| Listing 16.2.7-2.3 Adverse events of interest – Full Analysis Set | 439 |
| Listing 16.2.7-3.1 CV risk factors, Nilotinib exposure, glucose and total cholesterol rates for patients with cardiac and vascular adverse events of interest, Full Analysis Set | 440 |
| Listing 16.2.7-3.2 Cardiac and vascular adverse events of interest, Full Analysis Set | 441 |
| Listing 16.2.7-3.3 Outcomes and subsequent concomitant medications for patients with cardiac adverse events of interest, Full Analysis Set | 443 |
| Listing 16.2.7-3.4 Outcomes and subsequent concomitant medications for patients with vascular adverse events of interest, Full Analysis Set | 444 |
| Section 16.2.8 – Laboratory measurements | 445 |
| Listing 16.2.8-1.1 Hematology laboratory values and normal ranges – Full Analysis Set | 445 |
| Listing 16.2.8-2.1 Biochemistry laboratory values and normal ranges – Full Analysis Set | |
| Listing 16.2.8-3.1 Hematological data and molecular response in patients with absolute blasts higher than normal ranges, Full Analysis Set | 448 |
| Listing 16.2.8-3.2 Hematological data and molecular response in patients with absolute metamyelocytes higher than normal ranges, Full Analysis Set | 449 |
| Section 16.2.9 – Vital signs, physical findings and other observations related to safety listings | 450 |
| Listing 16.2.9-1.1 Vital signs – Full Analysis Set | 450 |
| Listing 16.2.9-2.1 Electrocardiograms – Full Analysis Set | 451 |
| Listing 16.2.9-2.2 Echocardiography – Full Analysis Set. | 451 |

| Listing 16.2.9-3.1 | Concomitant medications – Full Analysis Set | .452 |
|---|---|---|
| Listing 16.2.9- 3.2 | Prohibited concomitant medications – Full Analysis Set | .452 |
| Listing 16.2.9-4.1 | Prior Imatinib therapy– Full Analysis Set | .453 |
| • | Prior antineoplastic therapy, other than Imatinib – Full Analysis | |
| | Survival follow-up- Full Analysis set | |
| Listing 16.2.9-5.2 | Safety follow-up- Full Analysis set | .455 |
| Listing 16.2.9-6 | Prior imatinib exposure – LSC sub-study Full Analysis Set | .456 |

## 3. Shells and specification for CSR

## 3.1 Shells and specifications for sections 10 of the CSR (In-textText tables, listings and figures)

Document History – Changes compared to previous version of RAP module 7.1

- 1. General guidance
  - 1.1 Document headers
  - 1.2 Rules of presentation
  - 1.3 Document headers
  - 1.4 Presentation of table numbering and titles within this document
  - 1.5 Treatment group labels and ordering
  - 1.6 Distribution logistics
- 2. Overall table of contents for statistics and programming output

Tables, Listing Figures

- 3. Shells and specification for CSR
  - 3.1 Shells and specifications for sections 10 of the CSR (In-textText tables, listings and figures)

Section 10

- Table 10-1 Analysis sets All patients
- Table 10-2 Patient disposition during Induction/Consolidation phase and post-Randomization Consolidation phase -Enrolled patients
- Table 10-3 Demographic and characteristics at baseline Full Analysis Set
- Table 10-4 Disease history Full Analysis Set
- Table 10-5 Duration of exposure to study treatment during pre-randomization Induction/Consolidation Safety Set
- Table 10-6 Duration of exposure to study treatment during post-randomization Consolidation phase (ARM 2) - Subset of Safety Set randomized to Arm 2
- Table 11-1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase Full Analysis Set
- Table 11-2 Raw cumulative incidence of MR 4.0 during post-randomization consolidation phase (ARM 2) Subset of Full Analysis Set randomized to Arm 2
- Table 11-3 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase Full Analysis Set
- Table 11-4 Raw cumulative incidence of MR 4.5 during post-randomization consolidation phase (ARM 2) Subset of Full Analysis Set randomized to Arm 2
- Table 11-5 Primary endpoint, Molecular response MR4.0 at 12 months of TFR phase—Subset of Full Analysis Set entering the TFR phase
- Table 11-6 Secondary endpoint Kaplan-Meier analysis of treatment-free survival during the TFR phase Subset of Full Analysis Set entering the TFR phase

- Table 11-7 Secondary endpoint, Molecular response 4.0 during post-randomization consolidation phase (ARM 2) Subset of Full Analysis Set randomized to Arm 2
- Table 11-8 Secondary endpoint, Kaplan-Meier analysis of overall survival from Randomization–Randomized Set
- Table 12-1 Overall summary of treatment-emergent adverse events occurring during pre-randomization Induction/consolidation phase Full Analysis Set
- Table 12-2 Overall summary of treatment-emergent adverse events occurring during post-randomization consolidation phase (ARM 2) Subset of Full Analysis Set randomized to Arm 2
- Table 12-3 Overall summary of treatment-emergent adverse events occurring during re-treatment phase Subset of Full Analysis Set entering the re-treatment phase
- Table 12-4 Overall summary of adverse events occurring during TFR phase Subset of Full Analysis Set entering the TFR phase
- Table 12-5 Overall summary of frequent [1] treatment-emergent adverse events occurring during pre-randomization Induction/consolidation phase Full Analysis Set
- Table 12-6 Overall summary of frequent [1] treatment-emergent adverse events occurring during post-randomization Consolidation phase (ARM 2) Subset of Full Analysis Set randomized to Arm 2
- Table 12-7 Overall summary of frequent [1] treatment-emergent adverse events occurring during re-treatment phase Subset of Full Analysis Set entering the re-treatment phase
- Table 12-8 Overall summary of frequent [1] adverse events occurring during TFR phase Subset of Full Analysis Set entering the TFR phase
- Table 12-9 Serious treatment-emergent adverse events incidence, regardless of study drug relationship, by system organ class and preferred term during prerandomization Induction/consolidation phase overall and maximum grade 3/4 –Full Analysis Set
- Table 12-10 Serious treatment-emergent adverse events incidence, regardless of study drug relationship, by system organ class and preferred term during post-randomization consolidation phase (ARM 2) overall and maximum grade 3/4 Subset of Full Analysis Set randomized to Arm 2
- Table 12-11 Serious treatment-emergent adverse events incidence, regardless of study drug relationship, by system organ class and preferred term during retreatment phase overall and maximum grade 3/4 Subset of Full Analysis Set entering the re-treatment phase
- Table 12-12 Serious adverse events incidence, regardless of study drug relationship, by system organ class and preferred term during TFR phase overall and maximum grade 3/4 Subset of Full Analysis Set entering the TFR phase
- Table 12-13 Treatment-emergent adverse events of interest incidence, regardless of study drug relationship, by specific group and preferred term during Prerandomization Induction/consolidation phase –by treatment arm, overall and maximum grade 3/4 Full Analysis Set

- Table 12-14 Treatment-emergent adverse events of interest incidence by specific group and preferred term during post-randomization Consolidation phase (ARM 2) overall and maximum grade 3/4 Subset of Full Analysis Set randomized to Arm 2
- Table 12-15 Treatment-emergent adverse events of interest incidence by specific group and preferred term during re-treatment phase overall and maximum grade 3/4 Subset of Full Analysis Set entering the re-treatment phase
- Table 12-16 Adverse events of interest incidence by specific group and preferred term during TFR phase overall and maximum grade 3/4 Subset of Full Analysis Set entering the TFR phase
- Table 12-17 Treatment-emergent adverse events incidence leading to study drug discontinuation by system organ class and preferred term during prerandomization Induction/Consolidation phase overall and maximum grade 3/4 –Full Analysis Set
- Table 12-18 Treatment-emergent adverse events incidence leading to study drug discontinuation by system organ class and preferred term during post-randomizationphase (ARM 2) overall and maximum grade 3/4 Subset of Full Analysis Set randomized to Arm 2
- Table 12-19 On treatment deaths, by system organ class and preferred term during pre-randomization Induction/Consolidation phase Safety Set
- Table 12-20 On treatment deaths, by system organ class and preferred term during post-randomization consolidation phase (ARM 2) Subset of Safety Set randomized to Arm 2
- Table 12-21 On treatment deaths, by system organ class and preferred term during re-treatment phase Subset of Safety Set entering the re-treatment phase
- Listing 12-1 Listing of deaths Full Analysis Set
- Figure 11-1 Primary endpoint, Bar plot MR4.0 at 12 months of TFR phase –Subset of Full Analysis Set entering the TFR phase
- Figure 11-2 Kaplan-Meier analysis of treatment-free survival during the TFR phase –Subset of Full Analysis Set entering the TFR phase
- 3.2 Shells and specifications for Sections 14 and 16 of the CSR
- Section 14 tables, figures and graphs referred to but not included in the text
- Section 14.1 Demographic data
- Table 14.1-1.1 Enrollment by country and center All patients
- Table 14.1-1.2 Randomization by country and center Randomized patients
- Table 14.1-1.3 Patient disposition (Screening failures), All patients
- Table 14.1-2.1 Patient disposition during Induction/Consolidation phase and post-Randomization Consolidation phase -Enrolled patients
- Table 14.1-2.2 Patient disposition in each randomized arm Full Analysis Set
- Table 14.1-2.2.1 Patient disposition Enrolled patients in LSC substudy
- Table 14.1-2.3 Analysis sets –All patients
- Table 14.1-2.4 Not Randomized patients Enrolled patients
- Table 14.1-2.5 Patient disposition, Overall and by year-phase -Enrolled patients

- Table 14.1-2.6 Patients discontinued and reason for discontinuation Full Analysis Set
- Table 14.1-2.6.1 Patients discontinued and reason for discontinuation, SDV sensitivity Full Analysis Set
- Table 14.1-2.7 Summary of TFR phase Full Analysis Set
- Table 14.1-2.7.1 Summary of TFR phase, SDV sensitivity Full Analysis Set
- Table 14.1-2.8 Summary of re-treatment phase Full Analysis Set
- Table 14.1-2.8.1 Summary of re-treatment phase, SDV sensitivity Full Analysis Set
- Table 14.1-2.9 Summary of patients with relapse during the TFR phase but no entering re-treatment phase —Subset of Full Analysis Set entering the TFR phase
- Table 14.1-3.1 Demographic and characteristics at baseline–Full Analysis Set
- Table 14.1-3.1.1 Demographic and characteristics at baseline– LSC sub-study Full Analysis Set
- Table 14.1-4.1 Disease history Full Analysis Set
- Table 14.1-4.1.1 Disease history LSC sub-study Full Analysis Set
- Table 14.1-5.1 History of prior Imatinib therapy Full Analysis Set
- Table 14.1-5.1.1 History of prior Imatinib therapy LSC sub-study Full Analysis Set
- Table 14.1-5.2 Prior antineoplastic therapy, other than Imatinib, by ATC class and preferred term Full Analysis Set
- Table 14.1-6.1 Cardiovascular risk factors at baseline Full Analysis Set
- Table 14.1-6.2 Cardiovascular risk factors (based on medical history, laboratory values and vital signs at baseline) Full Analysis Set
- Section 14.2 Efficacy and other non-safety data (e.g. PK, PK/PD, Health Econ., QoL)
- Figure 14.2-1.1 Box-plot of BCR-ABL ratio (IS) during pre-randomization Induction/Consolidation phase Full Analysis Set
- Figure 14.2-1.2 Box-plot of BCR-ABL ratio (IS) during post-randomization Consolidation phase (ARM 2) – Subset of Full Analysis Set randomized to ARM 2
- Figure 14.2-1.3 Box-plot of BCR-ABL ratio (IS) during TFR phase Subset of Full Analysis Set entered TFR
- Figure 14.2-1.4 Box-plot of BCR-ABL ratio (IS) during re-treatment phase Subset of Full Analysis Set entered re-treatment
- Figure 14.2-1.5 Box-plot of BCR-ABL ratio (IS) during TFR phase , SDV sensitivity Subset of Full Analysis Set entered TFR
- Figure 14.2-1.6 Box-plot of BCR-ABL ratio (IS) during re-treatment phase, SDV sensitivity —Subset of Full Analysis Set entered re-treatment
- Figure 14.2-2.1.1 Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase Full Analysis Set

- Figure 14.2-2.1.2 Raw cumulative incidence of MMR during post-randomization Consolidation phase (ARM 2) Subset of Full Analysis Set randomized to ARM 2
- Figure 14.2-2.2.1 Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase by halving time of BCR-ABL (IS) ratio Full Analysis Set
- Figure 14.2-2.2.2 Raw cumulative incidence of MMR during post-randomization Consolidation phase (ARM 2) by halving time of BCR-ABL (IS) ratio Subset of Full Analysis Set randomized to ARM 2
- Figure 14.2-2.3.1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase Full Analysis Set
- Figure 14.2-2.3.2 Raw cumulative incidence of MR 4.0 during post-randomization Consolidation phase (ARM 2) Subset of Full Analysis Set randomized to ARM 2
- Figure 14.2-2.3.11 Raw cumulative incidence of MR 4.0, Randomized vs Not Randomized, during pre-randomization Induction/Consolidation phase Full Analysis Set
- Figure 14.2-2.4.1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase by halving time of BCR-ABL (IS) ratio Full Analysis Set
- Figure 14.2-2.4.2 Raw cumulative incidence of MR 4.0 during post-randomization Consolidation phase (ARM 2) by halving time of BCR-ABL (IS) ratio Subset of Full Analysis Set randomized to ARM 2
- Figure 14.2-2.5.1 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase Full Analysis Set
- Figure 14.2-2.5.11 Raw cumulative incidence of MR 4.5, Randomized vs Not Randomized, during pre-randomization Induction/Consolidation phase-Full Analysis Set
- Figure 14.2-2.5.2 Raw cumulative incidence of MR 4.5 during post-randomization Consolidation phase (ARM 2) Subset of Full Analysis Set randomized to ARM 2
- Figure 14.2-2.6.1 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase by halving time of BCR-ABL (IS) ratio Full Analysis Set
- Figure 14.2-2.6.2 Raw cumulative incidence of MR 4.5 during post-randomization Consolidation phase (ARM 2) by halving time of BCR-ABL (IS) ratio Subset of Full Analysis Set randomized to ARM 2
- Figure 14.2-2.7.1 Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase Full Analysis Set patients not reaching MMR at baseline
- Figure 14.2-2.8.1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase Full Analysis Set patients not reaching MR 4.0 at baseline
- Figure 14.2-2.9.1 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase Full Analysis Set patients not reaching MR 4.5 at baseline

- Figure 14.2-2.9.2 Raw cumulative incidence of MR 4.5 during post-randomization Induction/Consolidation phase (ARM 2)- Subset of Full Analysis Set patients not reaching MR 4.5 at baseline, randomized to ARM 2.
- Figure 14.2-2.10.1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase by BCR-ABL(IS) ratio at baseline Full Analysis Set
- Figure 14.2-2.10.2 Raw cumulative incidence of MR 4.0 during post-randomization Consolidation phase (ARM 2) by BCR-ABL(IS) ratio at baseline Subset of Full Analysis Set randomized to ARM 2.
- Figure 14.2-2.11.1 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase by BCR-ABL(IS) ratio at baseline Full Analysis Set
- Figure 14.2-2.11.2 Raw cumulative incidence of MR 4.5 during post-randomization Consolidation phase (ARM 2) by BCR-ABL(IS) ratio at baseline Subset of Full Analysis Set randomized to ARM 2.
- Figure 14.2-2.12.1 Box-plot of BCR-ABL ratio (IS) during pre-randomization Induction/Consolidation phase, excluding outliers (BCR-ABL (IS) ratio>10 Full Analysis Set
- Figure 14.2-2.12.2 Box-plot of BCR-ABL ratio (IS) over post-randomization Consolidation phase (ARM 2), excluding outliers (BCR-ABL (IS) ratio>10 Subset of Full Analysis Set randomized to ARM 2.
- Figure 14.2-13.1 Raw cumulative incidence of loss of MMR during TFR Subset of Full Analysis Set entering the TFR phase
- Figure 14.2-13.2 Raw cumulative incidence of MMR during re-treatment phase Subset of Full Analysis Set entering the re-treatment phase
- Figure 14.2-13.3 Raw cumulative incidence of loss of MMR during TFR, SDV sensitivity Subset of Full Analysis Set entering the TFR phase
- Figure 14.2-13.4 Raw cumulative incidence of MMR during re-treatment phase, SDV sensitivity Subset of Full Analysis Set entering the re-treatment phase
- Figure 14.2-14.1 Raw cumulative incidence of loss of MR4.0 during TFR phase Subset of Full Analysis Set entering the TFR phase
- Figure 14.2-14.2 Raw cumulative incidence of MR4.0 during re-treatment phase Subset of Full Analysis Set entering the re-treatment phase
- Figure 14.2-14.3 Raw cumulative incidence of loss of MR4.0 during TFR phase, SDV sensitivity –Subset of Full Analysis Set entering the TFR phase
- Figure 14.2-14.4 Raw cumulative incidence of MR4.0 during re-treatment phase, SDV sensitivity Subset of Full Analysis Set entering the re-treatment phase
- Figure 14.2-15.1 Raw cumulative incidence of loss of MR4.5 during TFR phase Subset of Full Analysis Set entering the TFR phase with MR4.5
- Figure 14.2-15.2 Raw cumulative incidence of MR4.5 during re-treatment phase Subset of Full Analysis Set entering the re-treatment phase
- Figure 14.2-15.3 Raw cumulative incidence of loss of MR4.5 during TFR phase, SDV sensitivity Subset of Full Analysis Set entering the TFR phase with MR4.5

- Figure 14.2-15.4 Raw cumulative incidence of MR4.5 during re-treatment phase, SDV sensitivity Subset of Full Analysis Set entering the re-treatment phase
- Figure 14.2-16 Bar plot MR4.0 at 12 months of TFR phase –Subset of Full Analysis Set entering the TFR phase
- Figure 14.2-16.2 Bar plot MR4.0 at month 12 TFR phase , SDV sensitivity –Subset of Full Analysis Set entering the TFR phase
- Figure 14.2-17.1 Kaplan-Meier analysis of progression-free survival during the TFR phase –Subset of Full Analysis Set entering the TFR phase
- Figure 14.2-17.2 Kaplan-Meier analysis of treatment-free survival during the TFR phase –Subset of Full Analysis Set entering the TFR phase
- Figure 14.2-17.3 Kaplan-Meier analysis of progression-free survival during the TFR phase, SDV sensitivity –Subset of Full Analysis Set entering the TFR phase
- Figure 14.2-17.4 Kaplan-Meier analysis of treatment-free survival during the TFR phase, SDV sensitivity –Subset of Full Analysis Set entering the TFR phase
- Figure 14.2-18.1 Kaplan-Meier analysis of reachievement of MMR, after loss of response in TFR –Subset of Full Analysis Set entering the re-treatment phase
- Figure 14.2-18.2 Kaplan-Meier analysis of reachievement of MR4.0, after loss of response in TFR Subset of Full Analysis Set entering the re-treatment phase
- Figure 14.2-18.3 Kaplan-Meier analysis of reachievement of MMR, after loss of response in TFR, SDV sensitivity –Subset of Full Analysis Set entering the re-treatment phase
- Figure 14.2-18.4 Kaplan-Meier analysis of reachievement of MR4.0, after loss of response in TFR, SDV sensitivity Subset of Full Analysis Set entering the re-treatment phase
- Table 14.2-1.1 Description of BCR-ABL (IS) ratio at Month 3 and halving time of BCR-ABL (IS) ratio subgroups Full Analysis Set
- Table 14.2-2.1.1 Molecular response MR4.0 at 12 months of TFR–Subset of Full Analysis Set entering the TFR phase
- Table 14.2-2.1.2 Molecular response MR4.0 at 12 months of TFR–Subset of Per Protocol Analysis Set entering the TFR phase
- Table 14.2-2.1.3 Molecular response MR4.0 at 12 months of TFR–Full Analysis Set
- Table 14.2-2.1.4 Molecular response MR4.0 at 12 months of TFR-Per Protocol Analysis Set
- Table 14.2-2.1.5 Molecular response MR4.0 at 12 months of TFR—Subset of Full Analysis Set entering the TFR phase with MR4.0 achieved up to month 3 of pre-randomization Induction/Consolidation phase
- Table 14.2-2.1.6 Molecular response MR4.0 at 12 months of TFR—Subset of Full Analysis Set entering the TFR phase with MR4.5 achieved up to month 3 of pre-randomization Induction/Consolidation phase
- Table 14.2-2.1.7 Molecular response MR4.0 at 12 months of TFR, SDV sensitivity Subset of Full Analysis Set entering the TFR phase
- Table 14.2-2.1.8 Molecular response MR4.0 at 12 months of TFR, SDV sensitivity Subset of Per Protocol Analysis Set entering the TFR phase

- Table 14.2-2.1.9 Molecular response MR4.0 at 12 months of TFR, SDV sensitivity Full Analysis Set
- Table 14.2-2.1.10 Molecular response MR4.0 at 12 months of TFR, SDV sensitivity

  —Per Protocol Analysis Set
- Table 14.2-2.2.1 Kaplan-Meier analysis of treatment-free survival during the TFR phase Subset of Full Analysis Set entering the TFR phase
- Table 14.2-2.2.2 Kaplan-Meier analysis of treatment-free survival during the TFR phase Subset of Per Protocol Analysis Set entering the TFR phase
- Table 14.2-2.2.3 Kaplan-Meier analysis of treatment-free survival during the TFR phase, SDV sensitivity Subset of Full Analysis Set entering the TFR phase
- Table 14.2-2.2.4 Kaplan-Meier analysis of treatment-free survival during the TFR phase, SDV sensitivity Subset of Per Protocol Analysis Set entering the TFR phase
- Table 14.2-2.3 Kaplan-Meier analysis of overall survival from Randomization—Randomized Set
- Table 14.2-2.4 Kaplan-Meier analysis of progression-free survival during the TFR phase Subset of Full Analysis Set entering the TFR phase
- Table 14.2-2.5 Kaplan-Meier analysis of overall survival from Randomization, SDV sensitivity –Randomized Set
- Table 14.2-2.6 Kaplan-Meier analysis of progression-free survival during the TFR phase, SDV sensitivity Subset of Full Analysis Set entering the TFR phase
- Table 14.2-3.1 Major molecular response during pre-randomization Induction/Consolidation phase –Full Analysis Set
- Table 14.2-3.1.1 Major molecular response during pre-randomization Induction/Consolidation phase LSC sub-study Full Analysis Set
- Table 14.2-3.2 Major molecular response during post-randomization consolidation phase (ARM 2)— Subset of Full Analysis Set randomized to Arm 2
- Table 14.2-3.2.1 Major molecular response during post-randomization consolidation phase (ARM 2) LSC sub-study Full Analysis Set randomized to Arm 2
- Table 14.2-3.3 Major molecular response during TFR phase –Subset of Full Analysis Set patients entered TFR phase
- Table 14.2-3.4 Major molecular response during re-treatment phase—Subset of Full Analysis Set patients entered re- treatment phase
- Table 14.2-3.5 Major molecular response during TFR phase –Subset of Full Analysis Set patients entered TFR phase with MR4.0 achieved up to month 3 of prerandomization Induction/Consolidation phase
- Table 14.2-3.6 Major molecular response during TFR phase –Subset of Full Analysis Set patients entered TFR phase with MR4.5 achieved up to month 3 of prerandomization Induction/Consolidation phase
- Table 14.2-3.7 Major molecular response during TFR phase, SDV sensitivity Subset of Full Analysis Set patients entered TFR phase
- Table 14.2-3.8 Major molecular response during re-treatment phase, SDV sensitivity

  —Subset of Full Analysis Set patients entered re- treatment phase

- Table 14.2-4.1 Molecular response 4.0 during pre-randomization Induction/Consolidation phase Full Analysis Set
- Table 14.2-4.1.1 Molecular response 4.0 during pre-randomization Induction/Consolidation phase LSC sub-study Full Analysis Set
- Table 14.2-4.2.1 Molecular response 4.0 during post-randomization consolidation phase (ARM 2) Subset of Full Analysis Set randomized to Arm 2
- Table 14.2-4.2.2 Molecular response 4.0 during post-randomization consolidation phase (ARM 2) Subset of Per Protocol randomized to Arm 2
- Table 14.2-4.2.11 Molecular response 4.0 during post-randomization consolidation phase (ARM 2) Subset of LSC sub-study Full Analysis Set randomized to Arm 2
- Table 14.2-4.3.1 Molecular response 4.0 during TFR phase Subset of Full Analysis Set entering the TFR phase
- Table 14.2-4.3.2 Molecular response 4.0 during TFR phase Subset of Per Protocol Analysis Set entering the TFR phase
- Table 14.2-4.3.3 Molecular response 4.0 during TFR phase, SDV sensitivity Subset of Full Analysis Set entering the TFR phase
- Table 14.2-4.4 Molecular response 4.0 during re-treatment phase Subset of Full Analysis Set entering the re-treatment phase
- Table 14.2-4.5 Molecular response 4.0 during TFR phase Subset of Full Analysis Set entering the TFR phase with MR4.0 achieved up to month 3 of prerandomization Induction/Consolidation phase
- Table 14.2-4.6 Molecular response 4.0 during TFR phase Subset of Full Analysis Set entering the TFR phase with MR4.5 achieved up to month 3 of prerandomization Induction/Consolidation phase
- Table 14.2-4.7 Molecular response 4.0 during re-treatment phase, SDV sensitivity Subset of Full Analysis Set entering the re-treatment phase
- Table 14.2-5.1 Molecular response 4.5 during pre-randomization Induction/Consolidation– Full Analysis Set
- Table 14.2-5.1.1 Molecular response 4.5 during pre-randomization Induction/Consolidation—LSC sub-study Full Analysis Set
- Table 14.2-5.2 Molecular response 4.5 during post-randomization consolidation phase (ARM 2) Subset of Full Analysis Set randomized to Arm 2
- Table 14.2-5.2.1 Molecular response 4.5 during post-randomization consolidation phase (ARM 2) Subset of LSC sub-study Full Analysis Set randomized to Arm 2
- Table 14.2-5.3 Molecular response 4.5 during TFR phase Subset of Full Analysis Set entering the TFR phase
- Table 14.2-5.4 Molecular response 4.5 during re-treatment phase Subset of Full Analysis Set entering the re-treatment phase
- Table 14.2-5.5 Molecular response 4.5 during TFR phase Subset of Full Analysis Set entering the TFR phase with MR4.0 achieved up to month 3 of prerandomization Induction/Consolidation phase

- Table 14.2-5.6 Molecular response 4.5 during TFR phase Subset of Full Analysis Set entering the TFR phase with MR4.5 achieved up to month 3 of prerandomization Induction/Consolidation phase
- Table 14.2-5.7 Molecular response 4.5 during TFR phase, SDV sensitivity Subset of Full Analysis Set entering the TFR phase
- Table 14.2-5.8 Molecular response 4.5 during re-treatment phase, SDV sensitivity Subset of Full Analysis Set entering the re-treatment phase
- Table 14.2-6.1 Raw cumulative incidence MMR during pre-randomization Induction/Consolidation phase Full Analysis Set
- Table 14.2-6.1.1 Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase LSC sub-study Full Analysis Set
- Table 14.2-6.2 Raw cumulative incidence MMR during post-randomization Consolidation phase (ARM 2) Subset of Full Analysis Set patients randomized to ARM 2
- Table 14.2-6.2.1 Raw cumulative incidence MMR during post-randomization Consolidation phase (ARM 2) - Subset of LSC sub-study Fulls Anslysis Set randomized to ARM 2
- Table 14.2-6.3 Raw cumulative incidence of MMR during re-treatment phase Subset of Full Analysis Set entering the re-treatment phase
- Table 14.2-6.4 Raw cumulative incidence of MMR during re-treatment phase, SDV sensitivity Subset of Full Analysis Set entering the re-treatment phase
- Table 14.2-7.1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase Full Analysis Set
- Table 14.2-7.1.1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase LSC sub-study Full Analysis Set
- Table 14.2-7.2 Raw cumulative incidence of MR 4.0 during post-randomization consolidation phase (ARM 2) Subset of Full Analysis Set randomized to ARM 2
- Table 14.2-7.2.1 Raw cumulative incidence of MR 4.0 during post-randomization consolidation phase (ARM 2) Subset of LSC sub-study Full Analysis Set randomized to ARM 2
- Table 14.2-7.3 Raw cumulative incidence of MR 4.0 during re-treatment phase Subset of Full Analysis Set entering the re-treatment phase
- Table 14.2-7.4 Raw cumulative incidence of MR 4.0 during re-treatment phase, SDV sensitivity Subset of Full Analysis Set entering the re-treatment phase
- Table 14.2-8.1 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase Full Analysis Set
- Table 14.2-8.1.1 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase LSC sub-study Full Analysis Set
- Table 14.2-8.2 Raw cumulative incidence of MR 4.5 during post-randomization consolidation phase (ARM 2) Subset of Full Analysis Set randomized to Arm 2
- Table 14.2-8.2.1 Raw cumulative incidence of MR 4.5 during post-randomization consolidation phase (ARM 2) Subset of LSC sub-study Full Analysis Set randomized to Arm 2

- Table 14.2-8.3 Raw cumulative incidence of MR 4.5 during re-treatment phase Subset of Full Analysis Set entering the re-treatment phase
- Table 14.2-8.4 Raw cumulative incidence of MR 4.5 during re-treatment phase, SDV sensitivity Subset of Full Analysis Set entering the re-treatment phase
- Table 14.2-9.1 Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase by halving time of BCR-ABL (IS) ratio Full Analysis Set
- Table 14.2-9.1.1 Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase by halving time of BCR-ABL (IS) ratio LSC sub-study Full Analysis Set
- Table 14.2-9.2 Raw cumulative incidence of MMR during post-randomization consolidation phase (ARM 2) by halving time of BCR-ABL (IS) ratio Subset of Full Analysis Set randomized to Arm 2
- Table 14.2-9.2.1 Raw cumulative incidence of MMR during post-randomization consolidation phase (ARM 2) by halving time of BCR-ABL (IS) ratio Subset of LSC sub-study Full Analysis Set randomized to Arm 2
- Table 14.2-9.3 Raw cumulative incidence of MMR during re-treatment phase by halving time of BCR-ABL (IS) ratio Subset of Full Analysis Set entering the re-treatment phase
- Table 14.2-10.1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase by halving time of BCR-ABL (IS) ratio Full Analysis Set
- Table 14.2-.10.1.1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase by halving time of BCR-ABL (IS) ratio LSC sub-study Full Analysis Set
- Table 14.2-10.2 Raw cumulative incidence of MR 4.0 during post-randomization consolidation phase (ARM 2) by halving time of BCR-ABL (IS) ratio Subset of Full Analysis Set randomized to Arm 2
- Table 14.2-10.2.1 Raw cumulative incidence of MR 4.0 during post-randomization consolidation phase (ARM 2) by halving time of BCR-ABL (IS) ratio Subset of LSC sub-study Full Analysis Set randomized to Arm 2
- Table 14.2-10.3 Raw cumulative incidence of MR4.0 during re-treatment phase by halving time of BCR-ABL (IS) ratio Subset of Full Analysis Set entering the re-treatment phase
- Table 14.2-11.1 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase by halving time of BCR-ABL (IS) ratio Full Analysis Set
- Table 14.2-.11.1.1 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase by halving time of BCR-ABL (IS) ratio LSC sub-study Full Analysis Set
- Table 14.2-11.2 Raw cumulative incidence of MR 4.5 during post-randomization consolidation phase (ARM 2) by halving time of BCR-ABL (IS) ratio Subset of Full Analysis Set randomized to Arm 2
- Table14.2-11.2.1 Raw cumulative incidence of MR 4.5 during post-randomization consolidation phase (ARM 2) by halving time of BCR-ABL (IS) ratio Subset of LSC sub-study Full Analysis Set randomized to Arm 2

- Table 14.2-11.3 Raw cumulative incidence of MR4.5 during re-treatment phase by halving time of BCR-ABL (IS) ratio Subset of Full Analysis Set entering the re-treatment phase
- Table 14.2-12.1 Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase by BCR-ABL (IS) ratio at Month 3 Full Analysis Set
- Table 14.2-12.1.1 Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase by BCR-ABL (IS) ratio at Month 3 LSC sub-study Full Analysis Set
- Table 14.2-12.2 Raw cumulative incidence of MMR during post-randomization consolidation phase (ARM 2) by BCR-ABL (IS) ratio at Month 3 Subset of Full Analysis Set randomized to Arm 2
- Table 14.2-12.2.1 Raw cumulative incidence of MMR during post-randomization consolidation phase (ARM 2) by BCR-ABL (IS) ratio at Month 3 Subset of LSC sub-study Full Analysis Set randomized to Arm 2
- Table 14.2-12.3 Raw cumulative incidence of MMR during re-treatment phase by BCR-ABL (IS) ratio at Month 3 Subset of Full Analysis Set entering the retreatment phase
- Table 14.2-13.1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase by BCR-ABL (IS) ratio at Month 3 Full Analysis Set
- Table 14.2-13.1.1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase by BCR-ABL (IS) ratio at Month 3 LSC sub-study Full Analysis Set
- Table 14.2-13.2 Raw cumulative incidence of MR 4.0 during post-randomization consolidation phase (ARM 2) by BCR-ABL (IS) ratio at Month 3 Subset of Full Analysis Set randomized to Arm 2
- Table 14.2-13.2.1 Raw cumulative incidence of MR 4.0 during post-randomization consolidation phase (ARM 2) by BCR-ABL (IS) ratio at Month 3 Subset of LSC sub-study Full Analysis Set randomized to Arm 2
- Table 14.2-13.3 Raw cumulative incidence of MR 4.0 during re-treatment phase by BCR-ABL (IS) ratio at Month 3 Subset of Full Analysis Set entering the retreatment phase
- Table 14.2-14.1 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase by BCR-ABL (IS) ratio at Month 3 Full Analysis Set
- Table 14.2-14.1.1 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase by BCR-ABL (IS) ratio at Month 3 LSC sub-study Full Analysis Set
- Table 14.2-14.2 Raw cumulative incidence of MR 4.5 during post-randomization consolidation phase (ARM 2) by BCR-ABL (IS) ratio at Month 3 Subset of Full Analysis Set randomized to Arm 2
- Table 14.2-14.2.1 Raw cumulative incidence of MR 4.5 during post-randomization consolidation phase (ARM 2) by BCR-ABL (IS) ratio at Month 3 Subset of LSC sub-study Full Analysis Set randomized to Arm 2

- Table 14.2-14.3 Raw cumulative incidence of MR 4.5 during re-treatment phase by BCR-ABL (IS) ratio at Month 3 Subset of Full Analysis Set entering the retreatment phase
- Table 14.2-15.1 Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase by Sokal Risk category– Full Analysis Set
- Table 14.2-15.2 Raw cumulative incidence of MR4.0 during pre-randomization Induction/Consolidation phase by Sokal Risk category—Full Analysis Set
- Table 14.2-15.3 Raw cumulative incidence of MR4.5 during pre-randomization Induction/Consolidation phase by Sokal Risk category—Full Analysis Set
- Table 14.2-16.1 Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase by time since initial diagnosis of CML–Full Analysis Set
- Table 14.2-16.2 Raw cumulative incidence of MR4.0 during pre-randomization Induction/Consolidation phase by time since initial diagnosis of CML Full Analysis Set
- Table 14.2-16.3 Raw cumulative incidence of MR4.5 during pre-randomization Induction/Consolidation phase by time since initial diagnosis of CML Full Analysis Set
- Table 14.2-17.1 Suboptimal response up to 24 months of pre-randomization Induction/Consolidation phase Full Analysis Set patients who prematurely discontinued the pre-randomization Induction/Consolidation phase
- Table 14.2-17.2 Suboptimal response up to 12 months of post-randomization Consolidation phase (ARM 2) Subset of Full Analysis Set patients who prematurely discontinued the Induction/Consolidation phase randomized to Arm 2
- Table 14.2-18.1 Suboptimal response up to 24 months of pre-randomization Induction/Consolidation phase Full Analysis Set
- Table 14.2-18.2 Suboptimal response up to 12 months of post-randomization Consolidation phase - Subset of Full Analysis Set, randomized to ARM 2
- Table 14.2-19.1 Kinetics of BCR-ABL (IS) ratio during pre-randomization Induction/Consolidation phase Full Analysis Set
- Table 14.2-19.1.1 Kinetics of BCR-ABL (IS) ratio during pre-randomization Induction/Consolidation phase LSC sub-study Full Analysis Set
- Table 14.2-19.2 Kinetics of BCR-ABL (IS) ratio during post-randomization consolidation phase (ARM 2) –Subset of Full Analysis Set randomized to Arm 2
- Table 14.2-19.2.1 Kinetics of BCR-ABL (IS) ratio during post-randomization consolidation phase (ARM 2) –Subset of LSC sub-study Full Analysis Set randomized to Arm 2
- Table 14.2-19.3 Kinetics of BCR-ABL (IS) ratio during TFR phase Subset of Full Analysis Set entering the TFR phase
- Table 14.2-19.4 Kinetics of BCR-ABL (IS) ratio during re-treatment phase Subset of Full Analysis Set entering the re-treatment phase
- Table 14.2-19.5 Kinetics of BCR-ABL (IS) ratio during TFR phase, SDV sensitivity

   Subset of Full Analysis Set entering the TFR phase

- Table 14.2-19.6 Kinetics of BCR-ABL (IS) ratio during re-treatment phase, SDV sensitivity Subset of Full Analysis Set entering the re-treatment phase
- Table 14.2-20.1 Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase Full Analysis Set patients not reaching MMR at baseline
- Table 14.2-20.2 Raw cumulative incidence of MMR during post-randomization Consolidation phase (ARM 2) Subset of Full Analysis Set patients not reaching MMR at baseline, randomized to ARM 2
- Table 14.2-21.1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase Full Analysis Set patients not reaching MR 4.0 at baseline
- Table 14.2-21.2 Raw cumulative incidence of MR 4.0 during post-randomization Consolidation phase (ARM 2) Subset of Full Analysis Set patients not reaching MR 4.0 at baseline, randomized to ARM 2
- Table 14.2-22.1 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase - Full Analysis Set patients not reaching MR 4.5 at baseline
- Table 14.2-22.2 Raw cumulative incidence of MR 4.5 during post-randomization Consolidation phase (ARM 2) Subset of Full Analysis Set patients not reaching MR 4.5 at baseline, randomized to ARM 2
- Table 14.2-22.3 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase Full Analysis Set patients not reaching MMR at baseline
- Table 14.2-22.4 Raw cumulative incidence of MR 4.0 during post-randomization Consolidation phase (ARM 2) Subset of Full Analysis Set patients not reaching MMR at baseline, randomized to ARM 2
- Table 14.2-22.5 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase Full Analysis Set patients not reaching MMR at baseline
- Table 14.2-22.6 Raw cumulative incidence of MR 4.5 during post-randomization Consolidation phase (ARM 2) Subset of Full Analysis Set patients not reaching MMR at baseline, randomized to ARM 2
- Table 14.2-23.1 Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase by BCR-ABL(IS) ratio at baseline Full Analysis Set
- Table 14.2-23.1.1 Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase by BCR-ABL (IS) ratio at baseline– LSC substudy Full Analysis Set
- Table 14.2-23.2 Raw cumulative incidence of MMR during post-randomization consolidation phase (ARM 2) by BCR-BL(IS) ratio at baseline Subset of Full Analysis Set, randomized to ARM 2
- Table 14.2-23.2.1 Raw cumulative incidence of MMR during post-randomization consolidation phase (ARM 2) by BCR-BL(IS) ratio at baseline Subset of LSC sub-study Full Analysis Set , randomized to ARM 2

- Table 14.2-23.3 Raw cumulative incidence of MMR during re-treatment phase by BCR-BL(IS) ratio at baseline Subset of Full Analysis Set entering the retreatment phase
- Table 14.2-24.1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase by BCR-ABL(IS) ratio at baseline Full Analysis Set
- Table 14.2-24.1.1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase by BCR-ABL (IS) ratio at baseline—LSC substudy Full Analysis Set
- Table 14.2-24.2 Raw cumulative incidence of MR 4.0 during post-randomization consolidation phase (ARM 2) by BCR-BL(IS) ratio at baseline Subset of Full Analysis Set, randomized to ARM 2
- Table 14.2-24.2.1 Raw cumulative incidence of MR 4.0 during post-randomization consolidation phase (ARM 2) by BCR-BL(IS) ratio at baseline Subset of LSC sub-study Full Analysis Set , randomized to ARM 2
- Table 14.2-24.3 Raw cumulative incidence of MR 4.0 during re-treatment phase by BCR-BL(IS) ratio at baseline Subset of Full Analysis Set entering the retreatment phase
- Table 14.2-25.1 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase by BCR-ABL(IS) ratio at baseline Full Analysis Set
- Table 14.2-25.1.1 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase by BCR-ABL (IS) ratio at baseline—LSC substudy Full Analysis Set
- Table 14.2-25.2 Raw cumulative incidence of MR 4.5 during post-randomization consolidation phase (ARM 2) by BCR-BL(IS) ratio at baseline Subset of Full Analysis Set, randomized to ARM 2
- Table 14.2-25.2.1 Raw cumulative incidence of MR 4.5 during post-randomization consolidation phase (ARM 2) by BCR-BL(IS) ratio at baseline Subset of LSC sub-study Full Analysis Set , randomized to ARM 2
- Table 14.2-25.3 Raw cumulative incidence of MR 4.5 during re-treatment phase by BCR-BL(IS) ratio at baseline Subset of Full Analysis Set entering the retreatment phase
- Table 14.2-26.1 Raw cumulative loss of MMR during TFR phase –Subset of Full Analysis Set entering the TFR phase
- Table 14.2-26.2 Raw cumulative loss of MR4.0 during TFR phase –Subset of Full Analysis Set entering the TFR phase
- Table 14.2-26.3 Raw cumulative loss of MR4.5 during TFR phase —Subset of Full Analysis Set entering the TFR phase with MR4.5
- Table 14.2-26.4 Raw cumulative loss of MMR during TFR phase, SDV sensitivity Subset of Full Analysis Set entering the TFR phase
- Table 14.2-26.5 Raw cumulative loss of MR4.0 during TFR phase, SDV sensitivity

  -Subset of Full Analysis Set entering the TFR phase
- Table 14.2-26.6 Raw cumulative loss of MR4.5 during TFR phase, SDV sensitivity
  —Subset of Full Analysis Set entering the TFR phase with MR4.5

- Table 14.2-27.1 Descriptive Statistics for CD34 cells: Total percentage LSC substudy Full Analysis Set
- Table 14.2-28.1 Descriptive Statistics for CD34+/CD38+ cells: Percentage from total CD34+ cells LSC sub-study Full Analysis Set
- Table 14.2-28.2 Descriptive Statistics for number of events sorted in CD34+/CD38+ cells LSC sub-study Full Analysis Set
- Table 14.2-28.3 Ph+ by HIS status, in CD34+/CD38+ cells LSC sub-study Full Analysis Set
- Table 14.2-28.4 Descriptive statistics of Ph+ in CD34+/CD38+ cells- LSC sub-study Full Analysis Set
- Table 14.2-28.5 BCR-ABL by RT-PCR status, in CD34+/CD38+ cells LSC substudy Full Analysis Set
- Table 14.2-29.1 Descriptive Statistics for CD34+/CD38- cells: Percentage from total CD34+ cells LSC sub-study Full Analysis Set
- Table 14.2-29.2 Descriptive Statistics for number of events sorted in CD34+/CD38-cells LSC sub-study Full Analysis Set
- Table 14.2-29.3 Ph+ by HIS status, in CD34+/CD38- cells LSC sub-study Full Analysis Set
- Table 14.2-29.4 Descriptive statistics of Ph+ in CD34+/CD38- cells- LSC sub-study Full Analysis Set
- Table 14.2-29.5 BCR-ABL by RT-PCR status, in CD34+/CD38- cells LSC substudy Full Analysis Set
- Table 14.2-30.1 Descriptive Statistics for Immunophenotypically aberrant CD34+ cells: Percentage from total CD34+ cells –LSC sub-study Full Analysis Set
- Table 14.2-30.2 Descriptive Statistics for number of events sorted in Immunophenotypically aberrant CD34+ cells LSC sub-study Full Analysis Set
- Table 14.2-30.3 Ph+ by HIS status, in Immunophenotypically aberrant CD34+ cells LSC sub-study Full Analysis Set
- Table 14.2-30.4 Descriptive statistics of Ph+ in Immunophenotypically aberrant CD34+ cells– LSC sub-study Full Analysis Set
- Table 14.2-30.5 BCR-ABL by RT-PCR status, in Immunophenotypically aberrant CD34+ cells LSC sub-study Full Analysis Set
- Table 14.2-31.1 Descriptive Statistics for Immunophenotypically aberrant CD34-cells: Percentage from total CD34+ cells LSC sub-study Full Analysis Set
- Table 14.2-31.2 Descriptive Statistics for number of events sorted in Immunophenotypically aberrant CD34- cells- LSC sub-study Full Analysis Set
- Table 14.2-31.3 Ph+ by HIS status, in Immunophenotypically aberrant CD34- cells LSC sub-study Full Analysis Set
- Table 14.2-31.4 Descriptive statistics of Ph+ in Immunophenotypically aberrant CD34- cells– LSC sub-study Full Analysis Set
- Table 14.2-31.5 BCR-ABL by RT-PCR status, in Immunophenotypically aberrant CD34- cells LSC sub-study Full Analysis Set

- Table 14.2-32.1 Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase by duration of prior exposure to Imatinib Full Analysis Set
- Table 14.2-32.1.1 Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase by prior Imatib treatment duration LSC sub-study Full Analysis Set
- Table 14.2-32.2 Raw cumulative incidence of MMR during post-randomization consolidation phase (ARM 2) by prior Imatib treatment duration Subset of Full Analysis Set, randomized to ARM 2
- Table 14.2-32.2.1 Raw cumulative incidence of MMR during post-randomization consolidation phase (ARM 2) by prior Imatib treatment duration Subset of LSC sub-study Full Analysis Set , randomized to ARM 2
- Table 14.2-32.3 Raw cumulative incidence of MMR during re-treatment phase by prior Imatib treatment duration Subset of Full Analysis Set entering the retreatment phase
- Table 14.2-33.1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase by prior Imatib treatment duration Full Analysis Set
- Table 14.2-33.1.1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase by prior Imatib treatment duration LSC substudy Full Analysis Set
- Table 14.2-33.2 Raw cumulative incidence of MR 4.0 during post-randomization consolidation phase (ARM 2) by prior Imatib treatment duration Subset of Full Analysis Set, randomized to ARM 2
- Table 14.2-33.2.1 Raw cumulative incidence of MR 4.0 during post-randomization consolidation phase (ARM 2) by prior Imatib treatment duration Subset of LSC sub-study Full Analysis Set , randomized to ARM 2
- Table 14.2-33.3 Raw cumulative incidence of MR 4.0 during re-treatment phase by prior Imatib treatment duration Subset of Full Analysis Set entering the retreatment phase
- Table 14.2-34.1 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase by prior Imatib treatment duration Full Analysis Set
- Table 14.2-34.1.1 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase by prior Imatib treatment duration LSC substudy Full Analysis Set
- Table 14.2-34.2 Raw cumulative incidence of MR 4.5 during post-randomization consolidation phase (ARM 2) by prior Imatib treatment duration Subset of Full Analysis Set, randomized to ARM 2
- Table 14.2-34.2.1 Raw cumulative incidence of MR 4.5 during post-randomization consolidation phase (ARM 2) by prior Imatib treatment duration Subset of LSC sub-study Full Analysis Set , randomized to ARM 2
- Table 14.2-34.3 Raw cumulative incidence of MR 4.5 during re-treatment phase by prior Imatib treatment duration Subset of Full Analysis Set entering the retreatment phase
- Section 14.3 Safety data

- Table 14.3-1.1 Duration of exposure to study treatment during pre-randomization Induction/Consolidation—Safety Set
- Table 14.3-1.1.1 Duration of exposure to study treatment during pre-randomization Induction/Consolidation—LSC sub-study Safety Set
- Table 14.3-1.2 Duration of exposure to study treatment during post-randomization Consolidation phase (ARM 2) - Subset of Safety Set randomized to Arm 2
- Table 14.3-1.2.1 Duration of exposure to study treatment during post-randomization Consolidation phase (ARM 2) Subset of LSC sub-study Safety Set randomized to Arm 2
- Table 14.3-1.1.3 Duration of exposure to study treatment during re-treatment phase Subset of Safety Set entering the re-treatment phase
- Table 14.3-1.1.21 Duration of exposure to study treatment during pre-randomization Induction/Consolidation phase, by stable MR4.0 at 24 months and halving time Safety Set
- Table 14.3-1.1.22 Duration of exposure to study treatment during pre-randomization Induction/Consolidation phase, by stable MR4.0 by 24 months and halving time Safety Set
- Table 14.3-2.1 Relative dose intensity and average daily dose during prerandomization Induction/Consolidation phase – Safety Set
- Table 14.3-2.1.1 Relative dose intensity and average daily dose during prerandomization Induction/Consolidation phase – LSC sub-study Safety Set
- Table 14.3-2.2 Relative dose intensity and average daily dose during post-randomization consolidation phase (ARM 2) Subset of Safety Set randomized to Arm 2
- Table 14.3-2.2.1 Relative dose intensity and average daily dose during post-randomization consolidation phase (ARM 2) Subset of LSC sub-study Safety Set randomized to Arm 2
- Table 14.3-2.3 Relative dose intensity and average daily dose during re-treatment phase Subset of Safety Set entering the re-treatment phase
- Table 14.3-3.1 Dose reduction and interruption during pre-randomization Induction/Consolidation phase Safety Set
- Table 14.3-3.1.1 Dose reduction and interruption during pre-randomization Induction/Consolidation phase LSC sub-study Safety Set
- Table 14.3-3.2 Dose reduction and interruption during post-randomization consolidation phase (ARM 2) Subset of Safety Set randomized to Arm 2
- Table 14.3-3.2.1 Dose reduction and interruption during post-randomization consolidation phase (ARM 2) Subset of LSC sub-study Safety Set randomized to Arm 2
- Table 14.3-3.3 Dose reduction and interruption during re-treatment phase Subset of Safety Set entering the re-treatment phase
- Table 14.3-4.1 Concomitant medication by ATC class and preferred term during prerandomization Induction/Consolidation phase Full Analysis Set
- Table 14.3-4.1.1 Concomitant medication by ATC class and preferred term during pre-randomization Induction/Consolidation phase LSC sub-study Full Analysis Set

- Table 14.3-4.2 Concomitant medication by ATC class and preferred term during post-randomization consolidation phase (ARM 2)— Subset of Full Analysis Set randomized to Arm 2
- Table 14.3-4.2.1 Concomitant medication by ATC class and preferred term during post-randomization consolidation phase (ARM 2)— Subset of LSC sub-study Full Analysis Set randomized to Arm 2
- Table 14.3-4.3 Concomitant medication by ATC class and preferred term during TFR phase Subset of Full Analysis Set entering the TFR phase
- Table 14.3-4.4 Concomitant medication by ATC class and preferred term during retreatment phase Subset of Full Analysis Set entering the re-treatment phase
- Table 14.3-5.1.1 Hematology shift table based on CTCAE grade during Pre-Randomization pre-randomization Induction/Consolidation –Full Analysis Set
- Table 14.3-5.1.2 Hematology shift table based on CTCAE grade during post-randomization consolidation phase (ARM 2)—Subset of Full Analysis Set randomized to Arm 2
- Table 14.3-5.1.3 Hematology shift table based on CTCAE grade during re-treatment phase Subset of Full Analysis Set entering the re-treatment phase
- Table 14.3-5.1.4 Hematology shift table based on CTCAE grade during whole study period Full Analysis Set
- Table 14.3-5.1.5 Hematology shift table based on CTCAE grade during re-treatment phase, SDV sensitivity Subset of Full Analysis Set entering the retreatment phase
- Table 14.3-5.1.6 Hematology shift table based on CTCAE grade during whole study period, SDV sensitivity–Full Analysis Set
- Table 14.3-5.2.1 Biochemistry shift table based on CTCAE grade during post-randomization consolidation phase (ARM 2)—Subset of Full Analysis Set randomized to Arm 2
- Table 14.3-5.2.2 Biochemistry shift table based on CTCAE grade during retreatment phase—Subset of Full Analysis Set entering the re-treatment phase
- Table 14.3-5.2.3 Biochemistry shift table based on CTCAE grade during whole study period Full Analysis Set
- Table 14.3-5.2.4 Biochemistry shift table based on CTCAE grade during retreatment phase, SDV sensitivity—Subset of Full Analysis Set entering the retreatment phase
- Table 14.3-5.2.5 Biochemistry shift table based on CTCAE grade during whole study period, SDV sensitivity Full Analysis Set
- Table 14.3-6.1.1 Hematology shift table based on normal range for parameters with no defined CTCAE grades during post-randomization consolidation phase (ARM 2)— Subset of Full Analysis Set randomized to Arm 2
- Table 14.3-6.1.2 Hematology shift table based on normal range for parameters with no defined CTCAE grades during re-treatment phase Subset of Full Analysis Set entering the re-treatment phase
- Table 14.3-6.1.3 Hematology shift table based on normal range for parameters with no defined CTCAE grades during whole study period –Full Analysis Set

- Table 14.3-6.1.4 Hematology shift table based on normal range for parameters with no defined CTCAE grades during re-treatment phase, SDV sensitivity Subset of Full Analysis Set entering the re-treatment phase
- Table 14.3-6.1.5 Hematology shift table based on normal range for parameters with no defined CTCAE grades during whole study period, SDV sensitivity –Full Analysis Set
- Table 14.3-6.2.1 Biochemistry shift table based on normal range for parameters with no defined CTCAE grades during post-randomization consolidation phase (ARM 2) Subset of Full Analysis Set randomized to Arm 2
- Table 14.3-6.2.2 Biochemistry shift table based on normal range for parameters with no defined CTCAE grades during re-treatment phase Subset of Full Analysis Set entering the re-treatment phase
- Table 14.3-6.2.3 Biochemistry shift table based on normal range for parameters with no defined CTCAE grades during whole study period –Full Analysis Set
- Table 14.3-6.2.4 Biochemistry shift table based on normal range for parameters with no defined CTCAE grades during re-treatment phase, SDV sensitivity Subset of Full Analysis Set entering the re-treatment phase
- Table 14.3-6.2.5 Biochemistry shift table based on normal range for parameters with no defined CTCAE grades during whole study period, SDV sensitivity –Full Analysis Set
- Table 14.3-7.1 ECG shift table based on notable values during Pre-randomization Induction Consolidation–Full Analysis Set
- Table 14.3-7.2 ECG shift table based on notable values during post-randomization consolidation phase (ARM 2) Subset of Full Analysis Set randomized to Arm 2
- Table 14.3-7.3 ECG shift table based on notable values during re-treatment phase Subset of Full Analysis Set entering the re-treatment phase
- Table 14.3-7.4 Notable ECG values during pre-randomization Ind/Cons –Full Analysis Set
- Table 14.3-7.5 Notable ECG values during post-randomization consolidation phase (ARM 2)— Subset of Full Analysis Set randomized to Arm 2
- Table 14.3-7.6 Notable ECG values during re-treatment phase Subset of Full Analysis Set entering the re-treatment phase
- Table 14.3-7.7 ECG shift table based on notable values during re-treatment phase, SDV sensitivity Subset of Full Analysis Set entering the re-treatment phase
- Table 14.3-7.8 Notable ECG values during re-treatment phase, SDV sensitivity Subset of Full Analysis Set entering the re-treatment phase
- Table 14.3-8.1 Echocardiography assessment at baseline Full Analysis Set
- Table 14.3-8.2 Echocardiography shift table based on overall interpretation Full Analysis Set
- Table 14.3-8.3 Echocardiography shift table based on overall interpretation, SDV sensitivity Full Analysis Set
- Table 14.3-9.1 Summary statistics of total cholesterol, HDL, LDL, glucose, microalbumin and HbA1c over Induction/Consolidation phase Full Analysis Set
- Table 14.3-9.2.1 Total cholesterol shift table based on specific levels during Induction Consolidation Full Analysis Set
- Table 14.3-9.2.2 Total cholesterol shift table based on specific levels during TFR phase Subset of Full Analysis Set entering the TFR phase
- Table 14.3-9.2.3 Total cholesterol shift table based on specific levels during Retreatment phase Subset of Full Analysis Set entering the Re-treatment phase
- Table 14.3-9.2.4 Total cholesterol shift table based on specific levels during TFR phase, SDV sensitivity Subset of Full Analysis Set entering the TFR phase
- Table 14.3-9.2.5 Total cholesterol shift table based on specific levels during Retreatment phase, SDV sensitivity Subset of Full Analysis Set entering the Re-treatment phase
- Table 14.3-10.1.1 Fasting glucose shift table based on specific levels during Induction Consolidation Full Analysis Set
- Table 14.3-10.1.2 Fasting glucose shift table based on specific levels during TFR phase Subset of Full Analysis Set entering the TFR phase
- Table 14.3-10.1.3 Fasting glucose shift table based on specific levels during Retreatment phase Subset of Full Analysis Set entering the Re-treatment phase
- Table 14.3-10.1.4 Fasting glucose shift table based on specific levels during TFR phase, SDV sensitivity Subset of Full Analysis Set entering the TFR phase
- Table 14.3-10.1.5 Fasting glucose shift table based on specific levels during Retreatment phase, SDV sensitivity Subset of Full Analysis Set entering the Re-treatment phase
- Table 14.3-11.1 Vital Signs during Induction Consolidation Full Analysis Set
- Table 14.3-11.2 Vital Signs during TFR phase Subset of Full Analysis Set entering the TFR phase
- Table 14.3-11.3 Vital Signs during Re-treatment phase Subset of Full Analysis Set entering the Re-treatment phase
- Table 14.3-11.4 Vital Signs during TFR phase, SDV sensitivity Subset of Full Analysis Set entering the TFR phase
- Table 14.3-11.5 Vital Signs during Re-treatment phase, SDV sensitivity Subset of Full Analysis Set entering the Re-treatment phase
- Table 14.3-12.1 Survival follow-up Full Analysis Set
- Table 14.3-12.2 Survival follow-up, SDV sensitivity Full Analysis Set
- Table 14.3-13.1 Safety follow-up Full analysis Set
- Table 14.3-13.2 Safety follow-up, SDV sensitivity Full analysis Set
- Section 14.3.1 Displays of adverse events
- Figure 14.3.1-1.1 Kaplan-Meier analysis of time-to-first CVEs during the prerandomization Induction/Consolidation phase – Full Analysis Set
- Figure 14.3.1-1.2 Kaplan-Meier analysis of time-to-first CVEs during the post-randomization consolidation phase (ARM 2) Subset of Full Analysis Set randomized to Arm 2

- Figure 14.3.1-1.3 Kaplan-Meier analysis of time-to-first CVEs during the TFR phase Subset of Full Analysis Set entering the TFR phase
- Figure 14.3.1-1.4 Kaplan-Meier analysis of time-to-first CVEs during the retreatment phase Subset of Full Analysis Set entering the re-treatment phase
- Figure 14.3.1-2.1 Number of sorted events by HIS CD34+/CD38+ cells
- Figure 14.3.1-2.2 Number of sorted events by PCR CD34+/CD38+ cells
- Figure 14.3.1-3.1 Number of sorted events by HIS CD34+/CD38- cells
- Figure 14.3.1-3.2 Number of sorted events by PCR CD34+/CD38- cells
- Figure 14.3.1-4.1 Number of sorted events by HIS Immunophenotypically aberrant CD34+ cells
- Figure 14.3.1-4.2 Number of sorted events by PCR Immunophenotypically aberrant CD34+ cells
- Figure 14.3.1-5.1 Number of sorted events by HIS Immunophenotypically aberrant CD34- cells
- Figure 14.3.1-5.2 Number of sorted events by PCR Immunophenotypically aberrant CD34- cells
- Figure 14.3.1-6.1 Number of HIS+ subjects CD34+/CD38+ cells LSC substudy Full Analysis Set
- Figure 14.3.1-6.2 Number of PCR subjects CD34+/CD38+ cells LSC substudy Full Analysis Set
- Figure 14.3.1-7.1 Number of HIS+ subjects CD34+/CD38- cells LSC substudy Full Analysis Set
- Figure 14.3.1-7.2 Number of PCR subjects CD34+/CD38- cells LSC substudy Full Analysis Set
- Figure 14.3.1-8.1 Number of HIS+ subjects Immunophenotypically aberrant CD34+ cells LSC substudy Full Analysis Set
- Figure 14.3.1-8.2 Number of PCR subjects Immunophenotypically aberrant CD34+ cells LSC substudy Full Analysis Set
- Figure 14.3.1-9.1 Number of HIS+ subjects Immunophenotypically aberrant CD34-cells LSC substudy Full Analysis Set
- Figure 14.3.1-9.2 Number of PCR subjects Immunophenotypically aberrant CD34-cells LSC substudy FAS
- Figure 14.3.1-10 Number of patients with detectable LSC LSC substudy Full Analysis Set
- Table 14.3.1-1.1 Overall summary of treatment-emergent adverse events occurring during pre-randomization Induction/consolidation phase Full Analysis Set
- Table 14.3.1-1.2 Overall summary of treatment-emergent adverse events occurring during post-randomization consolidation phase (ARM 2) Subset of Full Analysis Set randomized to Arm 2
- Table 14.3.1-1.3 Overall summary of treatment-emergent adverse events occurring during re-treatment phase Subset of Full Analysis Set entering the retreatment phase
- Table 14.3.1-1.4 Overall summary of adverse events occurring during TFR phase Subset of Full Analysis Set entering the TFR phase

- Table 14.3.1-2.1 Overall summary of frequent [1] treatment-emergent adverse events occurring during pre-randomization Induction/consolidation phase Full Analysis Set
- Table 14.3.1-2.2 Overall summary of frequent [1] treatment-emergent adverse events occurring during post-randomization consolidation phase (ARM 2) Subset of Full Analysis Set randomized to Arm 2
- Table 14.3.1-2.3 Overall summary of frequent [1] treatment-emergent adverse events occurring during re-treatment phase Subset of Full Analysis Set entering the re-treatment phase
- Table 14.3.1-2.4 Overall summary of frequent [1] adverse events occurring during TFR phase Subset of Full Analysis Set entering the TFR phase
- Table 14.3.1-3.1.1 Treatment Emergent adverse events incidence, regardless of study drug relationship, occurring during pre-randomization
  Induction/consolidation phase by system organ class and preferred term overall and maximum grade 3/4 Full Analysis Set
- Table 14.3.1-3.1.2 Treatment Emergent adverse events occurence, regardless of study drug relationship, occurring during pre-randomization Induction/consolidation phase by system organ class and preferred term overall and maximum grade 3/4 Full Analysis Set
- Table 14.3.1-3.2.1 Treatment Emergent adverse events incidence, regardless of study drug relationship, occurring during post-randomization consolidation phase (ARM 2) by system organ class and preferred term overall and maximum grade 3/4 Subset of Full Analysis Set randomized to Arm 2
- Table 14.3.1-3.2.2 Treatment Emergent adverse events occurence, regardless of study drug relationship, occurring during post-randomization consolidation phase (ARM 2) by system organ class and preferred term overall and maximum grade 3/4 Subset of Full Analysis Set randomized to Arm 2
- Table 14.3.1-3.3.1 Treatment-emergent adverse events incidence, regardless of study drug relationship, by system organ class and preferred term during retreatment phase overall and maximum grade 3/4 Subset of Full Analysis Set entering the re-treatment phase
- Table 14.3.1-3.3.2 Treatment-emergent adverse events occurrence, regardless of study drug relationship, by system organ class and preferred term during retreatment phase overall and maximum grade 3/4 Subset of Full Analysis Set entering the re-treatment phase
- Table 14.3.1-3.4.1 Adverse events incidence, regardless of study drug relationship, by system organ class and preferred term during TFR phase overall and maximum grade 3/4 Subset of Full Analysis Set entering the TFR phase
- Table 14.3.1-3.4.2 Adverse events occurrence, regardless of study drug relationship, by system organ class and preferred term during TFR phase overall and maximum grade 3/4 Subset of Full Analysis Set entering the TFR phase
- Table 14.3.1-3.5.1 Frequent [1] Treatment Emergent adverse events incidence, regardless of study drug relationship occurring during pre-randomization Induction/consolidation phase by system organ class and preferred term overall and maximum grade 3/4 Full Analysis Set

- Table 14.3.1-3.5.2 Frequent [1] Treatment Emergent adverse events incidence, regardless of study drug relationship occurring during post-randomization consolidation phase (ARM 2) by system organ class and preferred termoverall and maximum grade 3/4 Subset of Full Analysis Set randomized to Arm 2
- Table 14.3.1-3.5.3 Frequent [1] Treatment Emergent adverse events incidence, regardless of study drug relationship occurring during re-treatment phase by system organ class and preferred term- overall and maximum grade 3/4 Subset of Full Analysis Set entering the re-treatment phase
- Table 14.3.1-3.5.4 Frequent [1] adverse events incidence, regardless of study drug relationship occurring during TFR phase by system organ class and preferred term overall and maximum grade 3/4 Subset of Full Analysis Set entering the TFR phase
- Table 14.3.1-4.1.1 Serious treatment-emergent adverse events incidence, regardless of study drug relationship, by system organ class and preferred term during pre-randomization Induction/consolidation phase overall and maximum grade 3/4 –Full Analysis Set
- Table 14.3.1-4.1.2 Serious treatment-emergent adverse events occurence, regardless of study drug relationship, by system organ class and preferred term during pre-randomization Induction/consolidation phase overall and maximum grade 3/4 –Full Analysis Set
- Table 14.3.1-4.2.1 Serious treatment-emergent adverse events incidence, regardless of study drug relationship, by system organ class and preferred term during post-randomization consolidation phase (ARM 2) overall and maximum grade 3/4 Subset of Full Analysis Set randomized to Arm 2
- Table 14.3.1-4.2.2 Serious treatment-emergent adverse events occurrence, regardless of study drug relationship, by system organ class and preferred term during post-randomization consolidation phase (ARM 2) overall and maximum grade 3/4 Subset of Full Analysis Set randomized to Arm 2
- Table 14.3.1-4.3.1 Serious treatment-emergent adverse events incidence, regardless of study drug relationship, by system organ class and preferred term during re-treatment phase overall and maximum grade 3/4 Subset of Full Analysis Set entering the re-treatment phase
- Table 14.3.1-4.3.2 Serious treatment-emergent adverse events occurrence, regardless of study drug relationship, by system organ class and preferred term during re-treatment phase overall and maximum grade 3/4 Subset of Full Analysis Set entering the re-treatment phase
- Table 14.3.1-4.4.1 Serious adverse events incidence, regardless of study drug relationship, by system organ class and preferred term during TFR phase overall and maximum grade 3/4 Subset of Full Analysis Set entering the TFR phase
- Table 14.3.1-4.4.2 Serious adverse events occurence, regardless of study drug relationship, by system organ class and preferred term during TFR phase overall and maximum grade 3/4 Subset of Full Analysis Set entering the TFR phase
- Table 14.3.1-4.5.1 Frequent [1] Serious Treatment Emergent adverse events incidence, regardless of study drug relationship occurring during pre-

- randomization Induction/consolidation phase by system organ class and preferred term overall and maximum grade 3/4 Full Analysis Set
- Table 14.3.1-4.5.2 Frequent [1] Serious Treatment Emergent adverse events incidence, regardless of study drug relationship occurring during post-randomization consolidation phase (ARM 2) by system organ class and preferred term overall and maximum grade 3/4 Subset of Full Analysis Set randomized to Arm 2
- Table 14.3.1-4.5.3 Frequent [1] Serious Treatment Emergent adverse events incidence, regardless of study drug relationship occurring during re-treatment phase by system organ class and preferred term overall and maximum grade 3/4 Subset of Full Analysis Set entering the re-treatment phase
- Table 14.3.1-4.5.4 Frequent [1] Serious adverse events incidence, regardless of study drug relationship occurring during TFR phase by system organ class and preferred term overall and maximum grade 3/4 Subset of Full Analysis Set entering the TFR phase
- Table 14.3.1-4.6.1 Serious treatment-emergent adverse events incidence, suspected to be study drug related, by system organ class and preferred term during prerandomization Induction/consolidation phase overall and maximum grade 3/4 –Full Analysis Set
- Table 14.3.1-4.6.2 Serious treatment-emergent adverse events occurence, suspected to be study drug related, by system organ class and preferred term during prerandomization Induction/consolidation phase overall and maximum grade 3/4 –Full Analysis Set
- Table 14.3.1-4.7.1 Serious treatment-emergent adverse events incidence, suspected to be study drug related, by system organ class and preferred term during post-randomization consolidation phase (ARM 2) overall and maximum grade 3/4 Subset of Full Analysis Set randomized to Arm 2
- Table 14.3.1-4.7.2 Serious treatment-emergent adverse events occurrence, suspected to be study drug related, by system organ class and preferred term during post-randomization consolidation phase (ARM 2) overall and maximum grade 3/4 Subset of Full Analysis Set randomized to Arm 2
- Table 14.3.1-4.8.1 Serious treatment-emergent adverse events incidence, suspected to be study drug related, by system organ class and preferred term during retreatment phase overall and maximum grade 3/4 Subset of Full Analysis Set entering the re-treatment phase
- Table 14.3.1-4.8.2 Serious treatment-emergent adverse events occurrence, suspected to be study drug related, by system organ class and preferred term during retreatment phase overall and maximum grade 3/4 Subset of Full Analysis Set entering the re-treatment phase
- Table 14.3.1-4.9.1 Serious adverse events incidence, suspected to be study drug related, by system organ class and preferred term during TFR phase overall and maximum grade 3/4 Subset of Full Analysis Set entering the TFR phase
- Table 14.3.1-4.9.2 Serious adverse events occurrence, suspected to be study drug related, by system organ class and preferred term during TFR phase overall and maximum grade 3/4 Subset of Full Analysis Set entering the TFR phase

- Table 14.3.1-5.1.1 Treatment-emergent adverse events incidence leading to study drug discontinuation by system organ class and preferred term during prerandomization Induction/Consolidation phase overall and maximum grade 3/4 –Full Analysis Set
- Table 14.3.1-5.1.2 Treatment-emergent adverse events occurence leading to study drug discontinuation by system organ class and preferred term during prerandomization Induction/Consolidation phase overall and maximum grade 3/4 –Full Analysis Set
- Table 14.3.1-5.2.1 Treatment-emergent adverse events incidence leading to study drug discontinuation by system organ class and preferred term during post-randomization phase (ARM 2) overall and maximum grade 3/4 Subset of Full Analysis Set randomized to Arm 2
- Table 14.3.1-5.2.2 Treatment-emergent adverse events occurrence leading to study drug discontinuation by system organ class and preferred term during post-randomization phase (ARM 2)— overall and maximum grade 3/4 Subset of Full Analysis Set randomized to Arm 2
- Table 14.3.1-5.3.1 Treatment-emergent adverse events incidence leading to study drug discontinuation by system organ class and preferred term during retreatment phase overall and maximum grade 3/4 Subset of Full Analysis Set entering the re-treatment phase
- Table 14.3.1-5.3.2 Treatment-emergent adverse events occurrence leading to study drug discontinuation by system organ class and preferred term during retreatment phase overall and maximum grade 3/4 Subset of Full Analysis Set entering the re-treatment phase
- Table 14.3.1-6.1.1 Treatment-emergent adverse events incidence requiring dosage adjustment or temporarily interruption by system organ class and preferred term during pre-randomization Induction/ consolidation phase overall and maximum grade 3/4 —Full Analysis Set
- Table 14.3.1-6.1.2 Treatment-emergent adverse events occurrence requiring dosage adjustment or temporarily interruption by system organ class and preferred term during pre-randomization Induction/consolidation phase overall and maximum grade 3/4 –Full Analysis Set
- Table 14.3.1-6.2.1 Treatment-emergent adverse events incidence requiring dosage adjustment or temporarily interruption by system organ class and preferred term during post-randomization consolidation phase (ARM 2) overall and maximum grade 3/4 Subset of Full Analysis Set randomized to Arm 2
- Table 14.3.1-6.2.2 Treatment-emergent adverse events occurrence requiring dosage adjustment or temporarily interruption by system organ class and preferred term during post-randomization consolidation phase (ARM 2) overall and maximum grade 3/4 Subset of Full Analysis Set randomized to Arm 2
- Table 14.3.1-6.3.1 Treatment-emergent adverse events incidence requiring dosage adjustment or temporarily interruption by system organ class and preferred term during re-treatment phase overall and maximum grade 3/4 Subset of Full Analysis Set entering the re-treatment phase
- Table 14.3.1-6.3.2 Treatment-emergent adverse events occurrence requiring dosage adjustment or temporarily interruption by system organ class and preferred

- term during re-treatment phase overall and maximum grade 3/4 Subset of Full Analysis Set entering the re-treatment phase
- Table 14.3.1-6.4.1 Treatment-emergent adverse events of interest incidence, regardless of study drug relationship, by specific group and preferred term during Pre-randomization Induction/consolidation phase –by treatment arm, overall and maximum grade 3/4 Full Analysis Set
- Table 14.3.1-6.4.2 Treatment-emergent adverse events of interest occurrence, regardless of study drug relationship, by specific group and preferred term during Pre-randomization Induction/consolidation phase by treatment arm, overall and maximum grade 3/4 –Full Analysis Set
- Table 14.3.1-6.5.1 Treatment-emergent adverse events of interest incidence by specific group and preferred term during post-randomization consolidation phase (ARM 2) overall and maximum grade 3/4 Subset of Full Analysis Set randomized to Arm 2
- Table 14.3.1-6.5.2 Treatment-emergent adverse events of interest occurrence, by specific group and preferred term during post-randomization consolidation phase (ARM 2) overall and maximum grade 3/4 Subset of Full Analysis Set randomized to Arm 2
- Table 14.3.1-6.6.1 Treatment-emergent adverse events of interest incidence by specific group and preferred term during re-treatment phase overall and maximum grade 3/4 Subset of Full Analysis Set entering the re-treatment phase
- Table 14.3.1-6.6.2 Treatment-emergent adverse events of interest occurrence by specific group and preferred term during re-treatment phase overall and maximum grade 3/4 Subset of Full Analysis Set entering the re-treatment phase
- Table 14.3.1-6.7.1 Adverse events of interest incidence by specific group and preferred term during TFR phase overall and maximum grade 3/4 Subset of Full Analysis Set entering the TFR phase
- Table 14.3.1-6.7.2 Adverse events of interest occurrence by specific group and preferred term during TFR phase overall and maximum grade 3/4 Subset of Full Analysis Set entering the TFR phase
- Table 14.3.1-7.1.1 Treatment Emergent adverse events of interest incidence, regardless of study drug relationship, by specific group and preferred term and by cardiovascular risk factors during Pre-randomization Induction/consolidation phase by treatment arm, overall and maximum grade 3/4 Full Analysis Set
- Table 14.3.1-7.1.2 Treatment Emergent adverse events of interest occurrence, regardless of study drug relationship, by specific group and preferred term and by cardiovascular risk factors during Pre-randomization Induction/consolidation phase by treatment arm, overall and maximum grade 3/4 –Full Analysis Set
- Table 14.3.1-7.2.1 Treatment-emergent adverse events of interest incidence, regardless of study drug relationship, during post-randomization consolidation phase (ARM 2), by specific group and preferred term, and by cardiovascular risk factor—overall and maximum grade 3 or 4 Subset of Full Analysis Set randomized to Arm 2

- Table 14.3.1-7.2.2 Treatment-emergent adverse events of interest occurrence, regardless of study drug relationship, during post-randomization consolidation phase (ARM 2), by specific group and preferred term, and by cardiovascular risk factor overall and maximum grade 3 or 4 Subset of Full Analysis Set randomized to Arm 2
- Table 14.3.1-7.3.1 Treatment-emergent adverse events of interest incidence, regardless of study drug relationship, during re-treatment phase, by specific group and preferred term, and by cardiovascular risk factor Subset of Full Analysis Set entering the re-treatment phase
- Table 14.3.1-7.3.2 Treatment-emergent adverse events of interest occurrence, regardless of study drug relationship, during re-treatment phase, by specific group and preferred term, and by cardiovascular risk factor Subset of Full Analysis Set entering the re-treatment phase
- Table 14.3.1-7.4.1 Adverse events of interest incidence, regardless of study drug relationship, during TFR phase, by specific group and preferred term, and by cardiovascular risk factor Subset of Full Analysis Set entering the TFR phase
- Table 14.3.1-7.4.2 Adverse events of interest occurrence, regardless of study drug relationship, during TFR phase, by specific group and preferred term, and by cardiovascular risk factor Subset of Full Analysis Set entering the TFR phase
- Table 14.3.1-7.5.1 Treatment-emergent adverse events of interest incidence, regardless of study drug relationship, during pre-randomization Induction/consolidation phase, by specific group and preferred term and by 4 cardiovascular risk factors overall and maximum grade 3/4 –Full Analysis Set
- Table 14.3.1-7.5.2 Treatment-emergent adverse events of interest occurence, regardless of study drug relationship, during pre-randomization Induction/consolidation phase, by specific group and preferred term and by 4 cardiovascular risk factors overall and maximum grade 3/4 –Full Analysis Set
- Table 14.3.1-7.6.1 Treatment-emergent adverse events of interest incidence, regardless of study drug relationship, during post-randomization consolidation phase (ARM 2), by specific group and preferred term, and by 4 categories of cardiovascular risk factors— overall and maximum grade 3 or 4—Subset of Full Analysis Set randomized to Arm 2
- Table 14.3.1-7.6.2 Treatment-emergent adverse events of interest occurrence, regardless of study drug relationship, during post-randomization consolidation phase (ARM 2), by specific group and preferred term, and by 4 categories of cardiovascular risk factors overall and maximum grade 3 or 4 Subset of Full Analysis Set randomized to Arm 2
- Table 14.3.1-7.7.1 Treatment-emergent adverse events of interest incidence, regardless of study drug relationship, during re-treatment phase, by specific group and preferred term, and by 4 categories of cardiovascular risk factors Subset of Full Analysis Set entering the re-treatment phase
- Table 14.3.1-7.7.2 Treatment-emergent adverse events of interest occurrence, regardless of study drug relationship, during re-treatment phase, by specific

- group and preferred term, and by 4 categories of cardiovascular risk factors—Subset of Full Analysis Set entering the re-treatment phase
- Table 14.3.1-7.8.1 Adverse events of interest incidence, regardless of study drug relationship, during TFR phase, by specific group and preferred term, and by 4 categories of cardiovascular risk factors Subset of Full Analysis Set entering the TFR phase
- Table 14.3.1-7.8.2 Adverse events of interest occurrence, regardless of study drug relationship, during TFR phase, by specific group and preferred term, and by 4 categories of cardiovascular risk factors—Subset of Full Analysis Set entering the TFR phase
- Table 14.3.1-9.1 On treatment deaths, by system organ class and preferred term during pre-randomization Induction/Consolidation phase Safety Set
- Table 14.3.1-9.2 On treatment deaths, by system organ class and preferred term during post-randomization consolidation phase (ARM 2) Subset of Safety Set randomized to Arm 2
- Table 14.3.1-9.3 On treatment deaths, by system organ class and preferred term during re-treatment phase Subset of Safety Set entering the re-treatment phase
- Table 14.3.1-10.1.1 Cardiac and vascular adverse events of interest, incidence, by treatment arm during the pre-randomization induction/consolidation phase Full Analysis Set
- Table 14.3.1-10.1.2 Cardiac and vascular adverse events of interest, occurence, by treatment arm during the pre-randomization induction/consolidation phase Full Analysis Set
- Table 14.3.1-10.2.1 Cardiac and vascular adverse events of interest incidence, during the post-randomization consolidation phase (ARM 2) Subset of Full Analysis Set randomized to Arm 2
- Table 14.3.1-10.2.2 Cardiac and vascular adverse events of interest occurrence, during the post-randomization consolidation phase (ARM 2) Subset of Full Analysis Set randomized to Arm 2
- Table 14.3.1-10.3.1 Cardiac and vascular adverse events of interest, incidence, by treatment arm during the re-treatment phase Subset of Full Analysis Set entered re-treatment phase
- Table 14.3.1-10.3.2 Cardiac and vascular adverse events of interest, occurence, by treatment arm during the re-treatment phase Subset of Full Analysis Set entered re-treatment phase
- Table 14.3.1-10.4.1 Cardiac and vascular adverse events of interest, incidence, by treatment arm during the TFR phase Subset of Full Analysis Set entered TFR phase
- Table 14.3.1-10.4.2 Cardiac and vascular adverse events of interest, occurence, by treatment arm during the TFR phase Subset of Full Analysis Set entered TFR phase
- Table 14.3.1-10.5 Relationship between cardiac and vascular adverse events of interest with total cholesterol values Full Analysis Set
- Table 14.3.1-10.6 Relationship between cardiac and vascular adverse events of interest with glycemic values Full Analysis Set

- Table 14.3.1-11.1.1 Kaplan-Meier estimate of time-to-first CVEs during the prerandomization induction/consolidation phase – Full analysis set
- Table 14.3.1-11.1.2 Kaplan-Meier estimate of time-to-first CVEs during the post-randomization consolidation phase (ARM 2)—Subset of Full Analysis Set patients randomized on Arm 2
- Table 14.3.1-11.2 Kaplan-Meier estimate of time-to-first CVEs during the retreatment phase Subset of Full Analysis Set entering the re-treatment phase
- Table 14.3.1-12.1 Medical history by system organ class and preferred term- Full Analysis Set
- Table 14.3.1-13.1 Prior exposure to imatinib before screening, MMR, age, and Sokal by LSC detection category LSC sub-study Full Analysis Set
- Table 14.3.1-13.2.1 Percentage from total CD34+ cells, CD34+/CD38+ cells Subgroup of LSC sub-study Full Analysis Set, LSC detected
- Table 14.3.1-13.2.2 Percentage from total CD34+ cells, CD34+/CD38- cells Subgroup of LSC sub-study Full Analysis Set, LSC detected
- Table 14.3.1-13.2.3 Percentage from total CD34+ cells, Immunophenotypically aberrant CD34+ cells Subgroup of LSC sub-study Full Analysis Set, LSC detected
- Table 14.3.1-13.2.4 Percentage from total CD34+ cells, Immunophenotypically aberrant CD34 negative cells Subgroup of LSC sub-study Full Analysis Set, LSC detected
- Table 14.3.1-13.3.1 Percentage of Ph+ cells, CD34+/CD38- cells Subgroup of LSC sub-study Full Analysis Set, LSC detected
- Table 14.3.1-13.3.2 Percentage of Ph+ cells, CD34+/CD38- cells Subgroup of LSC sub-study Full Analysis Set, LSC detected
- Table 14.3.1-13.3.3 Percentage of Ph+ cells, Immunophenotypically aberrant CD34+ cells Subgroup of LSC sub-study Full Analysis Set, LSC detected
- Table 14.3.1-13.3.4 Percentage of Ph+ cells, Immunophenotypically aberrant CD34 negative cells Subgroup of LSC sub-study Full Analysis Set, LSC detected
- Table 14.3.1-13.4 Total Percentage of CD34+ cells- Subgroup of LSC sub-study Full Analysis Set, LSC detected
- Table 14.3.1-13.5 LSC detection LSC sub-study Full Analysis Set
- Section 14.3.2 Listings of deaths, other serious and significant adverse events
- Listing 14.3.2-1.1 Listing of deaths Full Analysis Set
- Listing 14.3.2-1.2 Listing of deaths SDV sensitivity Full Analysis Set
- Listing 14.3.2-2.1 Listing of adverse events of special interest Full Analysis Set
- Listing 14.3.2-2.2 Listing of adverse events leading to study drug discontinuation Full Analysis Set
- Listing 14.3.2-2.3 Listing of adverse events leading to study drug discontinuation during re-treatment phase Subset of Full Analysis Set entering the retreatment period
  - Section 14.3.3 Narratives of deaths, other serious and significant adverse events (non statistics and programming deliverables)
- Section 14.3.4 Abnormal laboratory value listings

- Listing 14.3.4-1.1 Listing of abnormal hematology laboratory value Full Analysis Set
- Listing 14.3.4-2.1 Listing of abnormal biochemistry laboratory value Full Analysis Set
- Section 16 Appendices
  - Section 16.1 Study information
  - Section 16.1.6 Listing of patients receiving test drug(s)/investigational product(s) from specific batches where more than one batch was used
  - Section 16.1.7 Randomization scheme and codes (subject identification and treatment assigned)
- Listing 16.1.7-1.1 Randomization schemes Randomized patients
  - Section 16.1.9 Documentation of statistical methods
- Listing 16.1.9.1 Raw Statistical output from Demographic and characteristics at baseline– Full Analysis Set
- Listing 16.1.9.1.1 Raw Statistical output from Demographic and characteristics at baseline– LSC sub-study Full Analysis Set
- Listing 16.1.9.2 Raw Statistical output from History of prior Imatinib therapy Full Analysis Set
- Listing 16.1.9.2.1 Raw Statistical output from History of prior Imatinib therapy LSC sub-study Full Analysis Set
- Listing 16.1.9.3 Raw Statistical output from Cardiovascular risk factors at baseline Full Analysis Set
- Listing 16.1.9.4.1 Raw Statistical output from Molecular response MR4.0 at 12 months of TFR–Subset of Full Analysis Set entering the TFR phase
- Listing 16.1.9.4.2 Raw Statistical output from Molecular response MR4.0 at 12 months of TFR–Subset of Per Protocol Analysis Set entering the TFR phase
- Listing 16.1.9.5.1 Raw Statistical output from Kaplan-Meier analysis of treatment-free survival during the TFR phase Subset of Full Analysis Set entering the TFR phase
- Listing 16.1.9.5.2 Raw Statistical output from Kaplan-Meier analysis of treatment-free survival during the TFR phase Subset of Per Protocol Analysis Set entering the TFR phase
- Listing 16.1.9.5.3 Raw Statistical output from Kaplan-Meier analysis of overall survival from Randomization–Randomized Set
- Listing 16.1.9.5.4 Raw Statistical output from Kaplan-Meier analysis of progression-free survival during the TFR phase Subset of Full Analysis Set entering the TFR phase
- Listing 16.1.9.6.1 Raw Statistical output from Kaplan-Meier estimate of time-to-first CVEs during the pre-randomization induction/consolidation phase Full analysis set
- Listing 16.1.9.6.2 Raw Statistical output from Kaplan-Meier estimate of time-to-first CVEs during the post-randomization consolidation phase (ARM 2)—Subset of Full Analysis Set patients randomized on Arm 2

- Listing 16.1.9.6.3 Raw Statistical output from Kaplan-Meier estimate of time-to-first CVEs during the re-treatment phase Subset of Full Analysis Set entering the re-treatment phase
- Section 16.2 Patient data listings
- Listing 16.2-1.1 Enrolled patients
- Section 16.2.1 Discontinued subjects
- Listing 16.2.1-1.1 Treatment and study completion Safety Set
- Listing 16.2.1-1.2 Study discontinuation Full Analysis Set
- Listing 16.2.1-1.3 Screen failures (All subjects enrolled)
- Section 16.2.2 Protocol deviations
- Listing 16.2.2-1.1 Protocol deviations Enrolled patients
- Section 16.2.3 Patients excluded from the efficacy analysis
- Listing 16.2.3-1.1 Analysis set All patients
- Section 16.2.4 Demographics and data at screening
- Listing 16.2.4-1.1 Demographic data Full Analysis Set
- Listing 16.2.4-2.1 Family history Full Analysis Set
- Listing 16.2.4-2.2 Disease history–Full Analysis Set
- Listing 16.2.4-3.1 Disease history I– Full Analysis Set
- Listing 16.2.4-3.2 Disease history II– Full Analysis Set
- Listing 16.2.4-3.3 Medical history/current medical condition Full Analysis Set
- Listing 16.2.4.4 Cardiovascular risk factors at baseline for patients with not evaluable CV risk factor, Full Analysis Set
- Section 16.2.5 Compliance and/or drug concentration data if available (including Bioanalytical Data Report)
- Listing 16.2.5-1.1 Dosage administration records Full Analysis Set
- Section 16.2.6 Individual efficacy response data
- Listing 16.2.6-1.1 BCR-ABL(IS) ratio and molecular responses during Induction/Consolidation and post-randomization consolidation phase (ARM 2) Full Analysis Set
- Listing 16.2.6-1.2 BCR-ABL(IS) ratio and molecular responses during TFR phase Subset of Full Analysis Set entering the TFR phase
- Listing 16.2.6-1.3 BCR-ABL(IS) ratio and molecular responses during re-treatment phase Subset of Full Analysis Set entering the re-treatment phase
- Listing 16.2.6-2.1 Criteria of successful TFR Subset of Full Analysis Set entering the TFR phase
- Listing 16.2.6-3.1 Assessment of progression-free survival during the TFR phase Subset of Full Analysis Set entering the TFR phase
- Listing 16.2.6-3.2 Assessment of treatment-free survival during the TFR phase Subset of Full Analysis Set entering the TFR phase
- Listing 16.2.6-3.3 Assessment of overall survival From Randomization Randomized set

- Listing 16.2.6-3.4 Assessment of relapse and treatment status during the TFR phase –Subset of Full Analysis Set entering the TFR phase and relapsed
- Listing 16.2.6-4.1 WBC and molecular response in patients with WBC increase (CTCAE grade>G1) Full Analysis Set
- Listing 16.2.6-5.1 Individual Efficacy data, Molecular response Full Analysis Set
- Listing 16.2.6-5.2 Individual Efficacy data, Bone-marrow I Full Analysis Set
- Listing 16.2.6-5.3 Individual Efficacy data, Bone -marrow II Full Analysis Set
- Listing 16.2.6-6.1.1 Total percentage of CD34+ cells LSC sub-study Full Analysis Set
- Listing 16.2.6-6.2.1 Percentage of cells from total CD34 positive—LSC sub-study Full Analysis Set
- Listing 16.2.6-6.3.1 Number of events sorted– LSC sub-study Full Analysis Set
- Listing 16.2.6-6.4.1 Ph+ by HIS- LSC sub-study Full Analysis Set
- Listing 16.2.6-6.5.1 BCR-ABL by RT-PCR-LSC sub-study Full Analysis Set
- Section 16.2.7 Adverse event listings
- Listing 16.2.7-1.1 All adverse events Full Analysis Set
- Listing 16.2.7-2.1 Serious adverse events Full Analysis Set
- Listing 16.2.7-2.2 Adverse events leading to study drug discontinuation Full Analysis Set
- Listing 16.2.7-2.3 Adverse events of interest Full Analysis Set
- Listing 16.2.7-3.1 CV risk factors, Nilotinib exposure, glucose and total cholesterol rates for patients with cardiac and vascular adverse events of interest, Full Analysis Set
- Listing 16.2.7-3.2 Cardiac and vascular adverse events of interest, Full Analysis Set
- Listing 16.2.7-3.3 Outcomes and subsequent concomitant medications for patients with cardiac adverse events of interest, Full Analysis Set
- Listing 16.2.7-3.4 Outcomes and subsequent concomitant medications for patients with vascular adverse events of interest, Full Analysis Set
- Section 16.2.8 Laboratory measurements
- Listing 16.2.8-1.1 Hematology laboratory values and normal ranges Full Analysis Set
- Listing 16.2.8-2.1 Biochemistry laboratory values and normal ranges Full Analysis Set
- Listing 16.2.8-3.1 Hematological data and molecular response in patients with absolute blasts higher than normal ranges, Full Analysis Set
- Listing 16.2.8-3.2 Hematological data and molecular response in patients with absolute metamyelocytes higher than normal ranges, Full Analysis Set
- Section 16.2.9 Vital signs, physical findings and other observations related to safety listings
- Listing 16.2.9-1.1 Vital signs Full Analysis Set
- Listing 16.2.9-2.1 Electrocardiograms Full Analysis Set
- Listing 16.2.9-2.2 Echocardiography Full Analysis Set

|-------------------------|--------------------|--------------|
| RAP Module 7.1 Addendum | 6-May-2021 (14:35) | CAMN107AIC05 |

| Listing 16.2.9-3.1 | Concomitant medications – Full Analysis Set |
|---|---|
| Listing 16.2.9- 3.2 | Prohibited concomitant medications – Full Analysis Set |
| Listing 16.2.9-4.1 | Prior Imatinib therapy– Full Analysis Set |
| Listing 16.2.9-4.2 | Prior antineoplastic therapy, other than Imatinib – Full Analysis |
| Set | |
| Listing 16.2.9-5.1 | Survival follow-up- Full Analysis set |
| Listing 16.2.9-5.2 | Safety follow-up- Full Analysis set |
| Listing 16.2.9-6 I | Prior imatinib exposure – LSC sub-study Full Analysis Set |

#### Table 10-1 Analysis sets - All patients

| Analysis set | All patients N=xx n (%) |
|----------------------------|-------------------------|
| Screened patients | xx (xx.x) |
| Screened successfully | xx (xx.x) |
| Re-screened | xx (xx.x) |
| Screen Failures | xx (xx.x) |
| Enrolled patients | xx (xx.x) |
| Randomized patients* | xx (xx.x) |
| Not Randomized patients | xx (xx.x) |
| Full Analysis Set (FAS)* | xx (xx.x) |
| Randomized patients* | xx (xx.x) |
| Not Randomized patients* | xx (xx.x) |
| Safety Set* | xx (xx.x) |
| Per Protocol Analysis Set* | xx (xx.x) |

<sup>-</sup> Randomized patients are all patients meeting eligibility criteria for randomization (i.e. achieved a sustained MR4.0 for at least 12 months in the Induction/Consolidation phase

of the study).

- Full Analysis Set (FAS) comprises all subjects who are enrolled, excluding patients with PD severity codes: 0, 8.

<sup>-</sup> Safety Set consists of all patients who received at least one dose of study drug, excluding patients with PD severity codes: 0, 5, 8.

- Per Protocol Analysis Set (PPS) comprises all subjects who are enrolled without major protocol

deviation (PD severity codes: 0, 1, 5, 8).
\* Patients without major PD.
Source: Post-text table 14.1-2.3

#### Table 10-2 Patient disposition during Induction/Consolidation phase and post-Randomization Consolidation phase -Enrolled patients

| Disposition<br>Reason | Arm 1<br>N=xx | N=xx | Total<br>N=xx |
|---|---|---|---|
| Patients enrolled | xx (xx.x) | | xx (xx.x) |
| Patients not-treated[1] | | | |
| Primary reason for study discontinuation | | | |
| Adverse event(s) Abnormal laboratory value(s) | xx (xx.x)<br>xx (xx.x) | | xx (xx.x)<br>xx (xx.x) |
| Abnormal test procedure result(s) | xx (xx.x) | | xx (xx.x) |
| Pregnancy<br>Protocol deviation<br>Subject withdrew consent | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) |
| Lost to follow-up<br>Administrative problems<br>Disease progression (CML) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) |
| Unstable MR4.0<br>New cancer (CML) therapy | xx (xx.x)<br>xx (xx.x) | | xx (xx.x)<br>xx (xx.x) |
| Relapse loss MMR/MR4<br>Other<br>Death | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) |
| Patients treated [2] Patients treated Discontinued from treatment | xx (xx.x)<br>xx (xx.x) | | xx (xx.x)<br>xx (xx.x) |
| Primary reason for study discontinuation | | | |
| Adverse event(s) Abnormal laboratory value(s) | xx (xx.x)<br>xx (xx.x) | | xx (xx.x)<br>xx (xx.x) |
| | • • • | | |

<sup>-</sup> Percentage is based on N.

reported as disc. Ind/Cons phase due to AE "Blast Crisis"- G2, should have Patient # been reported as disc. Ind/Cons phase due to Disease Progression, progression to Blast Crisis, as per Prot. Source: Post-text Table 14.1-2.1

<sup>[1]</sup> Patients who discontinued study after enrollment without taking study drug. [2] Patients who discontinued study during Induction/Consolidation phase.

<sup>- 15</sup> patients from ARM 2 discontinued during post-Randomization Consolidation phase.
- Patient # randomized to Arm 1 at and discontinued Ind/cons at - Patient # and discontinued Ind/cons at the same day for

Table 10-3 Demographic and characteristics at baseline – Full Analysis Set

| Characteristics at baseline | Arm 1<br>N=xx | N=xx | Total<br>N=xx | Comparison\$<br>p-value# |
|---|---|---|---|---|
| Age at baseline visit(Years) - n (%) < 65 >= 65 Missing | xx (xx.x)<br>xx (xx.x)<br>xx | | xx (xx.x)<br>xx (xx.x)<br>xx | 0.xxx |
| Age at baseline visit (Years) | | | | 0 |
| n<br>Mean<br>SD<br>25th Percentile<br>Median<br>75th Percentile<br>Min-Max | xxx<br>xx.x<br>xx.x<br>xx.x<br>xx.x<br>xx.x<br>xx.x | ••• | xxx<br>xx.x<br>x.xx<br>xx.x<br>xx.x<br>xx.x<br>xx.x | 0.xxx<br>0.xxx |
| Gender - n (%)<br>Female<br>Male<br>Missing | xx (xx.x)<br>xx (xx.x)<br>xx | ••• | xx (xx.x)<br>xx (xx.x)<br>xx | 0.xxx |
| <pre>If female, child bearing potential - n (%) Able to bear children Premenarche Post menopausal Sterile - of child bearing age Missing</pre> | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | 0.xxx |
| Race - n (%) Caucasian Black Asian Native American North African descent Unknown Other Missing | xx (xx.x) | | xx (xx.x) | 0.xxx |
| Body mass index (kg/m2) - n (%) Very severely underweight Severely underweight Underweight Normal Overweight Obese class I Obese class II Obese class III Missing | xx (xx.x) | | xx (xx.x) | 0.xxx |
| Body mass index (kg/m2)<br>n<br>Mean | xxx<br>xx.x | | xxx<br>xx.x | 0.xxx<br>0.xxx |

| Terri module /.1 mademadin | 0 111ay 2021 ( | 11.55) | | er min vi o / i me v |
|---|---|---|---|---|
| Characteristics at baseline | Arm 1<br>N=xx | N=xx | Total<br>N=xx | Comparison\$<br>p-value# |
| SD | x.xx | | X.XX | |
| 25th Percentile | XX.X | | XX.X | |
| Median | XX.X | | XX.X | |
| 75th Percentile | XX.X | | XX.X | |
| Min-Max | xx-xx | | xx-xx | |
| HIII HQX | AA AA | | AA AA | |
| ECOG performance | | | | |
| Status (WHO) - n (%) | | | | |
| 0 | xx (xx.x) | | xx (xx.x) | 0.xxx |
| 1 | xx (xx.x) | | xx (xx.x) | |
| 2 | xx (xx.x) | | xx (xx.x) | |
| 3 | xx (xx.x) | | xx (xx.x) | |
| 4 | xx (xx.x) | | xx (xx.x) | |
| Missing | XX (XX.X) | | XX (XX:X) | |
| 111331119 | ZZ | | AA | |
| Family history - n (%) | | | | |
| Diabetes | xx (xx.x) | | xx (xx.x) | |
| Hypertension | xx (xx.x) | | xx (xx.x) | |
| Dyslipidemia | xx (xx.x) | | xx (xx.x) | |
| Cardiac events | xx (xx.x) | | xx (xx.x) | |
| Cerebrovascular events | xx (xx.x) | | xx (xx.x) | |
| Peripheral arterial disease | xx (xx.x) | | xx (xx.x) | |
| Missing | XX | | XX | |
| 111551119 | 2121 | | 2121 | |
| Smoking history - n (%) | | | | |
| No | xx (xx.x) | | xx (xx.x) | 0.xxx |
| Yes | xx (xx.x) | | xx (xx.x) | V • |
| Ex-smoker | xx (xx.x) | | xx (xx.x) | |
| Missing | XX (XX.X) | ••• | XX (XX:X) | |
| 111001119 | | | | |
| If ex-smoker, time since | | | | |
| stopped smoking (months) | | | | |
| n | XXX | | XXX | 0.xxx |
| Mean | XX.X | | XX.X | 0.xxx |
| SD | X.XX | | X.XX | * |
| 25th Percentile | XX.X | | XX.X | |
| Median | XX.X | | XX.X | |
| 75th Percentile | XX.X | • • • | XX.X | |
| Min-Max | xx-xx | | xx-xx | |
| MIN MAX | AA AA | | AA AA | |
| If smoker or ex-smoker, use | | | | |
| of tobacco product in the | | | | |
| past month - n (%) | xx (xx.x) | | xx (xx.x) | |
| Cigarettes (including | xx (xx.x) | | xx (xx.x) | |
| roll-ups) | xx (xx.x) | | xx (xx.x) | |
| Cigars | xx (xx.x) | | xx (xx.x) | |
| Tobacco (e.g. pipe) | XX (XX•X) | | XX (XX.X) | |
| Others (e.g. pipe) | ΔΔ | | ΛΛ | |
| patches, chewing tobacco) | | | | |
| Missing | | | | |

<sup>-</sup> The last available assessment before or at date of start of study trt is taken as "baseline". BMI (kg/m2): very sev. underweight (< 15.0), sev. underweight (>=15.0-<=16.0), underweight (>16.0-<=18.5), normal (>18.5-<=25.0), overweight (>25.0-<=30.0), obese: class I (>30.0-<=35.0), class II (>35.0-<=40.0) and class III (over 40.0). Time since stopped smoking = (date of screen visit - date stopped smoking + 1) / 30.4375. Perc. based on the number of pat. Incl. in the analysis pop. (N). \$ Comparison Rand. vs Not Rand. # P-value: For cat. var. Pearson Chi-square or Fisher's exact test. For numeric var. independent t-test for means, Median test for medians. \* p-value<0.05, \*\* p-value<0.01.

Source: Post-text table: 14.1-3.1

#### Table 10-4 Disease history – Full Analysis Set

| Disease history | Arm 1<br>N=xx | <br>N=xx | Total<br>N=xx |
|---|---|---|---|
| | 14 222 | 11 2121 | 14 2121 |
| Time since initial diagnosis | | | |
| (months) | XXX | • • • | XXX |
| n<br>Maran | XX.X | | XX.X |
| Mean<br>SD | X.XX | | X.XX |
| 25th Percentile | XX.X<br>XX.X | | XX.X<br>XX.X |
| Median | XX.X | | XX.X |
| 75th Percentile | xx.x- xx.x | | XX.X- XX.X |
| Min-Max | | | |
| Time since initial diagnosis (years) | | | |
| - n (%)[1] | n=xx | | n=xx |
| <2 years | xx (xx.x) | | xx (xx.x) |
| 2 to 4 years | xx (xx.x) | | xx (xx.x) |
| 4 to 6 years | xx (xx.x) | | xx (xx.x) |
| 6 to 8 years | xx (xx.x) | | xx (xx.x) |
| 8 to 10 years | xx (xx.x) | | xx (xx.x) |
| 10 to 12 years | xx (xx.x) | | xx (xx.x) |
| >= 12 years | xx (xx.x) | | xx (xx.x) |
| Peripheral blood blasts % at | | • • • | |
| diagnosis | XXX | | XXX |
| n<br>Maan | XX.X | | XX.X |
| Mean<br>SD | X.XX | | x.xx<br>xx.x |
| 25th Percentile | XX.X<br>XX.X | | XX.X |
| Median | XX.X<br>XX.X | | XX.X |
| 75th Percentile | xx.x- xx.x | | xx.x- xx.x |
| Min-Max | AA.A AA.A | | 7V*V 7V*V |
| PB eosinophils % at diagnosis | | | |
| n | XXX | | XXX |
| Mean | XX.X | | XX.X |
| SD | X.XX | | X.XX |
| 25th Percentile | XX.X | | XX.X |
| Median | XX.X | | XX.X |
| 75th Percentile | XX.X | | XX.X |
| Min-Max | xx.x- xx.x | | xx.x- xx.x |
| PB basophils % at diagnosis | | | |
| n<br>Mean | XXX | • • • | XXX |
| SD SD | XX.X<br>X.XX | | XX.X<br>X.XX |
| 25th Percentile | XX.X | | XX.X |
| Median | XX.X | | XX.X |
| 75th Percentile | XX.X | | XX.X |
| Min-Max | xx.x- xx.x | | xx.x- xx.x |
| Platelets at diagnosis (10E9/L) | | | ******* |
| n | XXX | | XXX |
| Mean | XX.X | | XX.X |
| SD | X.XX | | X.XX |
| 25th Percentile | XX.X | | XX.X |
| Median | XX.X | | XX.X |
| 75th Percentile | XX.X | | XX.X |
| Min-Max | xx.x- xx.x | | xx.x- xx.x |
| Spleen size at diagnosis (cm under | | | |
| costal margin) | XXX | • • • | XXX |
| n<br>Maara | XX.X | | XX.X |
| Mean | X.XX | | X.XX |
| SD | XX.X | | XX.X |

| Novartis<br>AAP Module 7.1 Addendum | Confidential<br>6-May-2021 (14:35) | | Pag<br>CAMN107A |
|---|---|---|---|
| OF the Developed I. | | | |
| 25th Percentile | XX.X | | XX.X |
| Median | XX.X | | XX.X |
| 75th Percentile<br>Min-Max | xx.x- xx.x | | xx.x- xx.x |
| Extramedullary involvement other than hepato and/or splenomegaly | | | |
| - n (%)[1] | n=xx | | n=xx |
| Yes | xx (xx.x) | • • • | xx (xx.x) |
| No | xx (xx.x) | | xx (xx.x) |
| Sokal score | | | |
| n | xxx | | xxx |
| Mean | XX.X | | XX.X |
| SD | x.xx | | X.XX |
| 25th Percentile | XX.X | | XX.X |
| Median | XX.X<br>XX.X | | XX.X<br>XX.X |
| 75th Percentile | XX.X<br>XX.X | | XX.X<br>XX.X |
| Min-Max | | | |
| | xx.x- xx.x | | xx.x- xx.x |
| - n (%)[1] | n=xx | | U=XX |
| Low risk | xx (xx.x) | | xx (xx.x) |
| High risk | xx (xx.x) | | xx (xx.x) |
| Euro (Hasford) score | xxx | | xxx<br>xx.x<br>x.xx |
| Mean | XX.X | | XX.X |
| SD | X.XX | | XX.X |
| 25th Percentile | XX.X | | XX.X |
| Median | XX.X | | xx.x- xx.x |
| 75th Percentile | XX.X | | |
| Min-Max | xx.x- xx.x | | n=xx<br>xx (xx.x) |
| - n (%)[1] | 2-22 | | |
| | n=xx | • • • | xx (xx.x) |
| Low risk<br>Intermediate risk | xx (xx.x)<br>xx (xx.x) | | xx (xx.x) |
| High risk | xx (xx.x)<br>xx (xx.x) | | |
| EUTOS score | | | |
| n | XXX | | XXX |
| Mean | XX.X | | XX.X |
| SD | X.XX | | X.XX |
| 25th Percentile | XX.X | | XX.X |
| Median | XX.X | | XX.X |
| 75th Percentile | XX.X | | XX.X |
| Min-Max | xx.x- xx.x | | xx.x- xx.x |
| - n (%)[1] | n=xx | | n=xx |
| Low risk | xx (xx.x) | | xx (xx.x) |
| High risk | xx (xx.x) | | xx (xx.x) |
| Previous progression to AP/BC | n-vv | | 2-4 |
| - n (%)[1] | n=xx | • • • | N=XX |
| Yes<br>No | xx (xx.x)<br>xx (xx.x) | | xx (xx.x)<br>xx (xx.x) |
| Attempt to stop treatment with | | | |
| Imatinib | n=xx | | n=xx |
| - n (%)[1] | xx (xx.x) | - | xx (xx.x) |
| | xx (xx.x) | | xx (xx.x) |
| Yes | XX IXX.XI | | &X \ |

| Novartis RAP Module 7.1 Addendum | Confidential<br>6-May-2021 (14:35) | | Page 115<br>CAMN107AIC05 |
|---|---|---|---|
| BCR-ABL(IS) ratio at screening - n (%) [1] BCR-ABL(IS) > 1% BCR-ABL(IS) > 0.1% - <= 1% BCR-ABL(IS) > 0.01% - <= 0.1% BCR-ABL(IS) < -0.01% Undetectable BCR-ABL | n=xx<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | ••• | n=xx<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) |
| BCR-ABL(IS) ratio at Re-screening | g n=xx | | n=xx |
| - n (%)[1] BCR-ABL(IS) >1% | xx (xx.x)<br>xx (xx.x) | ••• | xx (xx.x)<br>xx (xx.x) |

<sup>-</sup> Time since initial diagnosis = (date of the baseline visit - date of initial diagnosis) /30.4375.

Source: Post-text table: 14.1-4.1

<sup>-</sup> Sokal score: low risk (<0.8), intermediate risk (>=0.8-<=1.2) and high risk (>1.2).

<sup>-</sup> Euro (Hasford) score: low risk (<=780), intermediate risk (>780-<=1480) and high risk (>1480).

<sup>-</sup> EUTOS score: low risk (<=87) and high risk (>87).

<sup>[1]</sup> Percentages over Number of non-missing.

Table 10-5 Duration of exposure to study treatment during pre-randomization Induction/Consolidation Safety Set

| | Arm 1<br>N=xx | Arm 2<br>N=xx | Randomized<br>N=xx | Not<br>Randomized<br>N=xx | Total<br>N=xx |
|---|---|---|---|---|---|
| Exposure (months) | | | | | |
| - n (%) | | | | | |
| < 6 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| >= 6 - < 12 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| >= 12 - < 18 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| >= 18 - < =24 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| > 24 | xx (xx.x) | | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Exposure (months) | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | X.XX | X.XX | X.XX | X.XX | X.XX |
| 25th Percentile | XX.X | XX.X | XX.X | XX.X | XX.X |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| 75th Percentile | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min-Max | xx.x- | xx.x- | xx.x- xx.x | xx.x- xx.x | xx.x- |
| | XX.X | XX.X | | | XX.X |

<sup>-</sup> Exposure (months) = (date of last administration - date of first administration in Induction/Consolidation phase + 1)/30.4375.

Source: Post-text table: 14.3-1.1

## Table 10-6 Duration of exposure to study treatment during post-randomization Consolidation phase (ARM 2) - Subset of Safety Set randomized to Arm 2

<< Programming note: Same shell as table 10-6.1 with arm 2 only.</pre>

Use <6, >=6 to <=12 and >12 categories.

Footnote:

Source: Post-text table: 14.3-1.2

<sup>-</sup> Safety Set consists of all patients who received at least one dose of study drug, excluding patients with PD severity codes (0, 5, 8).

<sup>-</sup> Exposure (months) = (date of last administration - date of first administration in post-randomization consolidation phase + 1)/30.4375.

<sup>-</sup> Safety Set consists of all patients who received at least one dose of study drug, excluding patients with PD severity codes (0, 5, 8).

Table 11-1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase – Full Analysis Set

| | Arm 1<br>N=xx | N=xx | Total<br>N=xx |
|---|---|---|---|
| Major molecular response at baseline<br>Number of responders | xx | | xx |
| Percentage (95% CI) | xx (xx.x, xx.x) | • • • | xx (xx.x, xx.x) |
| Cumulative major molecular response up to 3 months (Day 91) Cumulative number of responders | xx | | xx |
| Cumulative percentage (95% CI) | xx (xx.x, xx.x) | | xx (xx.x, xx.x) |
| Cumulative major molecular response up to 6 months (Day 183) Cumulative number of responders | xx | | xx |
| ••• | | | ••• |
| Cumulative major molecular response up to 9 months (Day 274) | | | |
| Cumulative major molecular response up to 12 months (Day 365) | ••• | | |
| Cumulative major molecular response up to 15 | ••• | | |
| months (Day 457) Cumulative major molecular response up to 18 | ••• | ••• | ••• |
| months (Day 548) Cumulative major molecular response up to2 | | • • • | |
| 21 months (Day 639) Cumulative Major molecular response up to 24 | | | |
| months (Day 731) | | | |

<sup>-</sup> Percentage based on the number of patients in the analysis population (N).

Source: Post-text table: 14.2-7.1

#### Table 11-2 Raw cumulative incidence of MR 4.0 during postrandomization consolidation phase (ARM 2) - Subset of Full Analysis Set randomized to Arm 2

<< Programming note: Same shell as table 11-1 for ARM 2 only>>

Source: Post-text table: 14.2-7.2

### Table 11-3 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase – Full Analysis Set

<< Programming note: Same shell as table 11-1 for MR4.5 >>

Source: Post-text table: 14.2-8.1

<sup>-</sup> Confidence interval calculated as per Clopper-Pearson exact method.

#### Table 11-4 Raw cumulative incidence of MR 4.5 during postrandomization consolidation phase (ARM 2) - Subset of Full Analysis Set randomized to Arm 2

<< Programming note: Same shell as table 11-2 for MR4.5 >>

Source: Post-text table: 14.2-8.2

### Table 11-5 Primary endpoint, Molecular response MR4.0 at 12 months of TFR phase–Subset of Full Analysis Set entering the TFR phase

| | Arm 1 | Arm 2 | Total |
|---|---|---|---|
| | N=xx | N=xx | N=xx |
| Number of responders | xx | xx | xx |
| Percentage (95% CI) | xx (xx.x, xx.x) | xx (xx.x, xx.x) | xx (xx.x, xx.x) |
| Comparison Arm 1 vs Arm 2 p-value\$ | 0.xxx* | | |

<sup>-</sup> Responders= Patients still in TFR with >=MR4.0, without molecular relapse.

Source: Post-text table: 14.2-2.1.1

<sup>-</sup> Confidence interval calculated as per Clopper-Pearson exact method.

<sup>-</sup> Percentage based on the number of patients included in the analysis population (N).

<sup>-</sup> Patients entered TFR considered for percentages denominator.

<sup>\$</sup> Pearson Chi-square test or Fisher's exact test depending on the crosstabulation frequencies. \* p-value<0.05, \*\* p-value<0.01.</pre>

Table 11-6 Secondary endpoint Kaplan-Meier analysis of treatment-free survival during the TFR phase – Subset of Full Analysis Set entering the TFR phase

| KM estimates | Arm 1 | Arm 2 |
|---|---|---|
| Number of patients - n(%) | | |
| with events | xx (xx.x) | xx (xx.x) |
| Relapse | xx (xx.x) | xx (xx.x) |
| Re-treatment with Nilotinib | xx (xx.x) | xx (xx.x) |
| Progression to AP-BC | xx (xx.x) | xx (xx.x) |
| Death from any cause | xx (xx.x) | xx (xx.x) |
| Relapse + Death from any | xx (xx.x) | xx (xx.x) |
| cause | | |
| | | occurring on the same date>> |
| with censorings | xx (xx.x) | xx (xx.x) |
| Time to event (months) | | |
| 25th percentile (95% CI) | xx (xx.x, xx.x) | xx (xx.x xx.x)) |
| Median (95% CI) | xx (xx.x xx.x)) | xx (xx.x xx.x)) |
| 75th percentile (95% CI) | xx (xx.x xx.x)) | xx (xx.x xx.x)) |
| Percentage of patients without | | |
| event - | | |
| Estimate n(%)(95% CI) | () ( | () () |
| 6 months | xx (xx.x) (xx.x, xx.x) | xx (xx.x) (xx.x, xx.x) |
| 12 months | xx (xx.x) (xx.x, xx.x) | xx (xx.x) (xx.x, xx.x) |
| 18 months | xx (xx.x) (xx.x, xx.x) | xx (xx.x) (xx.x, xx.x) |
| 24 months | xx (xx.x) (xx.x, xx.x) | xx (xx.x) (xx.x, xx.x) |
| 30 months | xx (xx.x) (xx.x, xx.x) | |
| 36 months | xx (xx.x) (xx.x, xx.x) | |

<sup>-</sup> NE: Not Estimable. Patients randomized to Arm 2 have a maximum of 24 months of TFR phase. - Event = first occurrence of relapse, re-treatment with nilotinib, progression to AP/BC or death for any cause. Censoring rule = patients who did not meet the event are censored at the first date occurring between: the last contact date, the end of TFR phase and the date of death. Time to event = (date of event - start date of TFR phase + 1)/30.4375.

Source: Post-text table:14.2-2.2.1

<sup>-</sup> n is the number of patients at risk at the timepoint (i.e. without event and still ongoing). The percentage of patients without event and the respective 95% C.I. are estimated from Kaplan Meier.

## Table 11-7 Secondary endpoint, Molecular response 4.0 during post-randomization consolidation phase (ARM 2) – Subset of Full Analysis Set randomized to Arm 2

| | Arm2<br>N=xx |
|---|---|
| Rate of major molecular response at<br>Baseline<br>Number of responders<br>Response Rate % (95% CI) | xx<br>xx (xx.x, xx.x) |
| Rate of major molecular response at<br>Month 27<br>Number of responders<br>Response Rate % (95% CI) | xx<br>xx (xx.x, xx.x) |
| Rate of major molecular response at<br>Month 27 (Nominal visit*)<br>Number of responders<br>Response Rate % (95% CI) | xx<br>xx (xx.x, xx.x) |
| Rate of major molecular response at Month 30 | |
| Rate of major molecular response at Month 33 | |
| Rate of major molecular response at Month 36 | |
| Rate of major molecular response at Month 36 (Nominal vist*) | |

<sup>-</sup> Rate was computed using time-window as described in the RAP Module 3.

#### << Programming note:

-The number of responders at Month  $\mathbf x$  is obtained by counting all patients with a response on the last assessment of time-window  $\mathbf x$ .

-The percentage is obtained by dividing the number of responders by N.>>

Source: Post-text table:14.2-4.2.1

<sup>-</sup> Percentage based on the number of patients included in the analysis population  $(\mathbf{N})$  .

<sup>-</sup> Confidence interval calculated as per Clopper-Pearson exact method.

 $<sup>\</sup>mbox{*}$  Nominal visit is according to the CRF record, regardless of time-window derived visit.

#### Table 11-8 Secondary endpoint, Kaplan-Meier analysis of overall survival from Randomization–Randomized Set

| KM estimates | Arm 1 | Arm 2 |
|---|---|---|
| Number of patients - n(%) | | |
| with events (deaths) | xx (xx.x) | xx (xx.x) |
| with censorings | xx (xx.x) | xx (xx.x) |
| Time to event (months) | | |
| 25th percentile (95% CI) | xx (xx.x, xx.x) | xx (xx.x xx.x)) |
| Median (95% CI) | xx (xx.x xx.x)) | xx (xx.x xx.x)) |
| 75th percentile (95% CI) | xx (xx.x xx.x)) | xx (xx.x xx.x)) |
| Percentage of patients without | | |
| event - | | |
| Estimate n(%)(95% CI) 6 months | vv (vv v) (vv v vv v) | xx (xx.x) (xx.x, xx.x) |
| 12 months | xx (xx.x) (xx.x, xx.x) | |
| 18 months | xx (xx.x) (xx.x, xx.x) | |
| 24 months | xx (xx.x) (xx.x, xx.x) | |
| 30 months | xx (xx.x) (xx.x, xx.x) | , , , ,,, |
| 36 months | xx (xx.x) (xx.x, xx.x) | |

<sup>-</sup> NE: Not Estimable. Event = death for any cause.

Source: Post-text table:14.2-2.3

<sup>-</sup> Censoring rule = patients who did not meet the event are censored at the first date occurring between:

the last contact date and the date of death.

<sup>-</sup> Time to event = (date of event - Randomization date + 1)/30.4375.

<sup>-</sup> n is the number of patients at risk at the timepoint (i.e. without event and still ongoing)

<sup>-</sup> The percentage of patients without event and the respective 95% C.I. are estimated from Kaplan Meier.

Table 12-1 Overall summary of treatment-emergent adverse events occurring during pre-randomization Induction/consolidation phase – Full Analysis Set

| Adverse event category | Arm 1<br>N=xx | N=XX | Total<br>N=xx |
|---|---|---|---|
| Any adverse events | xx (xx.x) | | xx (xx.x) |
| Any AE of special interest | xx (xx.x) | | xx (xx.x) |
| Grading of AEs NCI-CTCAE Grade 4 NCI-CTCAE Grade 3 NCI-CTCAE Grade 2 NCI-CTCAE Grade 1 NCI-CTCAE Missing | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) |
| Death | xx (xx.x) | | xx (xx.x) |
| AEs suspected to be related to nilotinib | xx (xx.x) | | xx (xx.x) |
| AEs leading to study drug discontinuation | xx (xx.x) | | xx (xx.x) |
| AEs requiring dosage adjustment or temporarily interruption | xx (xx.x) | • • • | xx (xx.x) |
| Serious AEs | xx (xx.x) | | xx (xx.x) |
| Serious AEs suspected to be related to nilotinib | xx (xx.x) | • • • | xx (xx.x) |
| Serious AEs leading to study drug discontinuation | xx (xx.x) | • • • | xx (xx.x) |

<sup>-</sup> For patient # due to reconciliation discrepancies, safety database reported AE term "Endometriosis" as a SAE, while in clinical database this AE was not recorded as an SAE.

- Only TEAEs from pre-rand. Ind./Cons. phase have been included. A pat. with mult. occur. of an AE is counted only once in the AE categ.; Perc. based on the pop. number (N). AESI CVEs (IHD), CVEs (PAOD), CVEs (ICD) and CVEs (others) were based on grouped MedDRA terms as descr. in the CRS. Treatment Arm 1/Arm 2: 24/36 months, Re-treatment max Arm 1/Arm 2: 36/24 months. Patient # rep. as disc. Ind/Cons phase due to AE "Blast Crisis"-G2, should have been reported as disc. Ind/Cons due to Dis. progr. to Blast Crisis, as per Prot. For pat. # AE "PHLEGMON FOOT - BIG TOE RIGHT" is rep. as PT "Cellulitis" in the AE list. and as PT "Osteoarthritis" in the SAE list. PT for the same AE has been wrongly dec. and reconc. was not req. a perfect match of the PT. Source: Post-text table: 14.3.1-1.1

# Table 12-2 Overall summary of treatment-emergent adverse events occurring during post-randomization consolidation phase (ARM 2) – Subset of Full Analysis Set randomized to Arm 2

| Adverse event category | Arm2<br>N=xx |
|---|---|
| Any adverse events | xx (xx.x) |
| Any AE of special interest | xx (xx.x) |
| Grading of AEs NCI-CTCAE Grade 4 NCI-CTCAE Grade 3 NCI-CTCAE Grade 2 NCI-CTCAE Grade 1 NCI-CTCAE Missing | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) |
| Death | xx (xx.x) |
| AEs suspected to be related to nilotinib | xx (xx.x) |
| AEs leading to study drug discontinuation | xx (xx.x) |
| AEs requiring dosage adjustment or temporarily interruption | xx (xx.x) |
| Serious AEs | xx (xx.x) |
| Serious AEs suspected to be related to nilotinib | xx (xx.x) |
| Serious AEs leading to study drug discontinuation | xx (xx.x) |

<sup>-</sup> Only treatment emergent adverse events from post-randomization consolidation phase are included in this table. A patient with multiple occurrences of an AE is counted only once in the AE category. Percentage based on the population number (N). AE of special interest CVEs (IHD), CVEs (PAOD), CVEs (ICD) and CVEs (others) are based on grouped MedDRA terms as described in the Case Retrieval Sheet.

Source: Post-text table: 14.3.1-1.2

<sup>-</sup> Patients randomized to Arm 2 have 12 months of treatment post-randomization and a maximum of 24 months of re-treatment.

Table 12-3 Overall summary of treatment-emergent adverse events occurring during re-treatment phase – Subset of Full Analysis Set entering the re-treatment phase

| Adverse event category | Arm 1 | Arm 2 | Total |
|---|---|---|---|
| | N=xx | N=xx | N=xx |
| Any adverse events | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any AE of special interest | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Grading of AEs | | | |
| NCI-CTCAE Grade 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| NCI-CTCAE Grade 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| NCI-CTCAE Grade 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| NCI-CTCAE Grade 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| NCI-CTCAE Missing | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Death | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AEs suspected to be related to nilotinib | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AEs leading to study drug discontinuation | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AEs requiring dosage adjustment or temporarily interruption | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Serious AEs | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Serious AEs suspected to be related to nilotinib | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Serious AEs leading to study drug discontinuation | xx (xx.x) | xx (xx.x) | xx (xx.x) |

<sup>-</sup> Only treatment emergent adverse events from re-treatment phase are included in this table. A patient with multiple occurrences of an AE is counted only once in the AE category. Percentage based on the population number (N). AE of special interest CVEs (IHD), CVEs (PAOD), CVEs (ICD) and CVEs (others) are based on grouped MedDRA terms as described in the Case Retrieval Sheet. - Patients randomized to Arm 1 have 24 months of treatment and a maximum of 36 months of retreatment. Patients randomized to Arm 2 have 36 months of treatment and a maximum of 24 months of re-treatment.

Source: Post-text table: 14.3.1-1.3


CAMN107AIC05

| Adverse event category | Arm 1<br>N=xx | Arm 2<br>N=xx | Total<br>N=xx |
|---|---|---|---|
| Any adverse events | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any AE of special interest | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Grading of AEs | | | |
| NCI-CTCAE Grade 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| NCI-CTCAE Grade 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| NCI-CTCAE Grade 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| NCI-CTCAE Grade 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| NCI-CTCAE Missing | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Death | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AEs suspected to be related to nilotinib | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AE occurring within 30 days after TFR end | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AE occurring after 30 days after TFR end | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Serious AEs | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Serious AEs suspected to be related to nilotinib | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Source: Post-text table: 14.3.1-1.4

Only adverse events from TFR phase are included in this table.A patient with multiple occurrences of an AE is counted only once in the AE category. Percentage based on the population number (N). Patients randomized to Arm 1 have 24 months of treatment and a maximum of 36 months of re-treatment. Patients randomized to Arm 2 have 36 months of treatment and a maximum of 24 months of re-treatment. AE of special interest CVEs (IHD), CVEs (PAOD), CVEs (ICD) and CVEs (others) are based on grouped MedDRA terms as described in the Case Retrieval Sheet.

## Table 12-5 Overall summary of frequent [1] treatment-emergent adverse events occurring during pre-randomization Induction/consolidation phase – Full Analysis Set

<< Programming note: Same shell as table 12-1 using the following footnotes:

Source: Post-text table: 14.3.1-2.1 [1] Frequent AE defined as an AE present at 5% or more for at least one treatment Arm. Only treatment emergent adverse events from pre-rand. ind./cons. phase are included in this table. A patient with multiple occurrences of an AE is counted only once in the AE category. Percentage based on the population number (N). AE of special interest CVEs (IHD), CVEs (PAOD), CVEs (ICD) and CVEs (others) are based on grouped MedDRA terms as described in the Case Retrieval Sheet.

- Treatment Arm 1/Arm 2: 24/36 months, Re-treatment max Arm 1/Arm 2: 36/24 months. Source: Post-text table: 14.3.1-2.1

# Table 12-6 Overall summary of frequent [1] treatment-emergent adverse events occurring during post-randomization Consolidation phase (ARM 2) – Subset of Full Analysis Set randomized to Arm 2

<< Programming note: Same shell as table 12-2 adding the following footnote:
[1] Frequent AE defined as an AE present at 5% or more of the ARM2 patients.
Source: Post-text table: 14.3.1-2.2</pre>

## Table 12-7 Overall summary of frequent [1] treatment-emergent adverse events occurring during re-treatment phase – Subset of Full Analysis Set entering the re-treatment phase

<< Programming note: Same shell as table 12-3 adding the following footnote:
 [1] Frequent AE defined as an AE present at 5% or more for at least one treatment
Arm.</pre>

Source: Post-text table: 14.3.1-2.3

## Table 12-8 Overall summary of frequent [1] adverse events occurring during TFR phase – Subset of Full Analysis Set entering the TFR phase

<< Programming note: Same shell as table 12-4 adding the following footnote:</pre>

[1] Frequent AE defined as an AE present at 5% or more for at least one treatment Arm.

Source: Post-text table: 14.3.1-2.4

Table 12-9 Serious treatment-emergent adverse events incidence, regardless of study drug relationship, by system organ class and preferred term during pre-randomization Induction/consolidation phase - overall and maximum grade 3/4 -Full Analysis Set


| | Arr<br>N=2 | • | Total | | | |
|---|---|---|---|---|---|---|
| Primary system<br>organ class<br>Preferred term | All<br>grades<br>n (%) | Grade<br>3/4<br>n (%) | | | All<br>grades<br>n (%) | Grade<br>3/4<br>n (%) |
| Any Primary<br>system organ<br>class | xx (xx.x) | xx (xx.x) | ••• | ••• | xx (xx.x) | xx (xx.x) |
| Cardiac<br>disorders | xx (xx.x) | xx (xx.x) | | | xx (xx.x) | xx (xx.x) |
| Angina pectoris | xx (xx.x) | xx (xx.x) | | | xx (xx.x) | xx (xx.x) |
| Bradycardia NOS | xx (xx.x) | xx (xx.x) | | | xx (xx.x) | xx (xx.x) |
| Oedema NOS | xx (xx.x) | xx (xx.x) | | | xx (xx.x) | xx (xx.x) |
| Tachycardia NOS | xx (xx.x) | xx (xx.x) | • • • | • • • | xx (xx.x) | xx (xx.x) |

- For patient # \_\_\_\_\_, due to reconciliation discrepancies, safety database reported AE term "Endometriosis" as a SAE, while in clinical - For patient # database this AE was not recorded as an SAE.

<sup>-</sup> Only TEAEs from pre-rand. Ind./Cons. phase have been included. Primary SOC presented alphab.; PTs are sorted within prim. SOC in desc. freq. of 'All grades' column. Perc. based on pop. number (N). Treatment Arm 1/Arm 2: 24/36 months, Re-trt max Arm 1/Arm 2: 36/24 months. A pat. with mult. occur. of an AE is counted only once in the AE cat.; A pat. with mult. AEs within a prim. SOC is counted only once in the total row. AEs occur. more than 30 days after last study trt. exp. date are not summarized. For pat. # AE "PHLEGMON FOOT - BIG TOE RIGHT" is rep. as PT "Cellulitis" in the AE list. and as PT "Osteoarthritis" in the SAE listing. PT for the same AE has been wrongly dec. and reconc. was not req. a perfect match of the PT. Source: Post-text table 14.3.1-4.1.1

Table 12-10 Serious treatment-emergent adverse events incidence, regardless of study drug relationship, by system organ class and preferred term during post-randomization consolidation phase (ARM 2) – overall and maximum grade 3/4 – Subset of Full Analysis Set randomized to Arm 2

| | Arm2 | |
|--------------------------------|------------|-----------|
| | N=xxx | |
| Primary system organ class | All grades | Grade 3/4 |
| Preferred term | n (%) | n (%) |
| Any primary system organ class | xx (xx.x) | xx (xx.x) |
| Cardiac disorders | xx (xx.x) | xx (xx.x) |
| Angina pectoris | xx (xx.x) | xx (xx.x) |
| Bradycardia NOS | xx (xx.x) | xx (xx.x) |
| Oedema NOS | xx (xx.x) | xx (xx.x) |
| Tachycardia NOS | xx (xx.x) | xx (xx.x) |
| etc. | | |

<sup>-</sup> Only treatment emergent adverse events from post-rand. cons. phase (ARM 2) are included in this table. Primary system organ classes are presented alphabetically; preferred terms are sorted within primary system organ class in descending frequency of 'All grades' column. Percentage based on the number of patients included in the analysis population (N).

Source: Post-text table: 14.3.1-4.2.1

Table 12-11 Serious treatment-emergent adverse events incidence, regardless of study drug relationship, by system organ class and preferred term during re-treatment phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the re-treatment phase

<< Programming note: Same shell as table 12.9 for re-treatment period>>
Source: Post-text table: 14.3.1-4.3.1

Table 12-12 Serious adverse events incidence, regardless of study drug relationship, by system organ class and preferred term during TFR phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the TFR phase

<< Programming note: Same shell as table 12.9 for TFR and replacing 1st footnote:
- Only adverse events from TFR phase are included in this table.>>

Source: Post-text table: 14.3.1-4.4.1

<sup>-</sup> Treatment post-randomization Arm 2: 12 months, Re-treatment max Arm 2: 24 months.

<sup>-</sup> A patient with multiple occurrences of an AE is counted only once in the AE category.

<sup>-</sup> A patient with multiple adverse events within a primary system organ class is counted only once in the total row. Adverse events occurring more than 30 days after last study treatment exposure date are not summarized.

Table 12-13 Treatment-emergent adverse events of interest incidence, regardless of study drug relationship, by specific group and preferred term during Pre-randomization Induction/consolidation phase –by treatment arm, overall and maximum grade 3/4 – Full Analysis Set

| | Arı<br>N= | n 1<br>xxx | | ··· | | tal<br>xxx |
|---|---|---|---|---|---|---|
| Specific group<br>Preferred term | All<br>grades<br>n (%) | Grade<br>3/4<br>n (%) | Grade<br>3/4<br>n (%) | All<br>grades<br>n (%) | Grade<br>3/4<br>n (%) | All<br>grades<br>n (%) |
| All AESI | xx (xx.x) | xx (xx.x) | | | xx (xx.x) | xx (xx.x) |
| Group 1<br>PT1<br>PT2 | xx (xx.x)<br>xx (xx.x) | , , | | | xx (xx.x)<br>xx (xx.x) | |
| Group 2<br>PT1<br>PT2 | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | | | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) |

<sup>-</sup> Only TEAEs from pre-rand. ind./cons. phase have been incl. in this table. Specific groupings are pres. alphabetically; PTs are sorted within each group in desc. frequency of 'All grades' column. Perc. based on the pop. number (N). Trt Arm 1/Arm 2: 24/36 months, Re-trt max Arm 1/Arm 2: 36/24 months. A patient with mult. occurrences of an AE is counted only once in the AE category. A patient with mult. AEs within a group is counted only once in the total row. AESI: CVEs (IHD), CVEs (PAOD), CVEs (ICD) and CVEs (others) are based on grouped MedDRA terms as described in the Case Retrieval Sheet. AEs occurring more than 30 days after last study treatment exposure date are not summarized.

Source: Post-text table: 14.3.1-6.4.1

Table 12-14 Treatment-emergent adverse events of interest incidence by specific group and preferred term during post-randomization Consolidation phase (ARM 2) - overall and maximum grade 3/4 -Subset of Full Analysis Set randomized to Arm 2

| Specific group Preferred term | Arm2<br>N=xx | |
|-------------------------------|--------------|-----------|
| | All grades | Grade 3/4 |
| | n (%) | n (%) |
| All AESI | xx (xx.x) | xx (xx.x) |
| Group 1 | | |
| PT 1 | xx (xx.x) | xx (xx.x) |
| PT 2 | xx (xx.x) | xx (xx.x) |
| ect | xx (xx.x) | xx (xx.x) |
| Group 2 | | |
| PT 1 | xx (xx.x) | xx (xx.x) |
| PT 2 | xx (xx.x) | xx (xx.x) |
| ect | xx (xx.x) | xx (xx.x) |
| ect | | |

<sup>-</sup> Only TEAEs from post-rand. cons. phase incl. in this table. Specific groups are pres. alphabetically; PTs are sorted within each group in desc. frequency of 'All grades' column. Perc. based on the number of patients included in the analysis pop. (N). Trt post-rand. Arm 2: 12 months, Re-trt max Arm 2: 24 months. A pat. with mult. occurrences of an AE is counted only once in the AE category. A pat. with mult. AEs within a group is counted only once in the total row. AESI:CVEs (IHD), CVEs (PAOD), CVEs (ICD) and CVEs (others) are based on grouped MedDRA terms as described in the Case Retrieval Sheet. AEs occurring more than 30 days after last study trt exp. date are not summarized. Source: Post-text table: 14.3.1-6.5.1
# Table 12-15 Treatment-emergent adverse events of interest incidence by specific group and preferred term during re-treatment phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the re-treatment phase

| Specific<br>group<br>Preferred | Arm<br>N=3 | | Arm<br>N=: | | Total<br>N=xx | |
|---|---|---|---|---|---|---|
| term | All grades n (%) | Grade 3/4<br>n (%) | All grades n (%) | Grade 3/4<br>n (%) | All grades<br>n (%) | Grade 3/4<br>n (%) |
| All AESI | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Group 1 | | | | | | |
| PT 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ect | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Group 2 | | | | | | |
| PT 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ect | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ect | | | | | | |

<sup>-</sup> Only TEAEs from re-trt phase are included in this table. Specific groups are alph. presented; PTs are sorted within each group in desc. freq. of 'All grades' column. Perc. based on the number of pat. included in the analysis pop. (N). Trt Arm 1/Arm 2: 24/36 months, Re-trt max Arm 1/Arm 2: 36/24 months. A patient with mult. occurrences of an AE is counted only once in the AE category. A patient with mult. AEs within a group is counted only once in the total row. AE of special interest CVEs (IHD), CVEs (PAOD), CVEs (ICD) and CVEs (others) are based on grouped MedDRA terms as described in the Case Retrieval Sheet.AEs occurring more than 30 days after last study trt exp. date are not summarized. Source: Post-text table: 14.3.1-6.6.1

# Table 12-16 Adverse events of interest incidence by specific group and preferred term during TFR phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the TFR phase

<< Programming note: Same shell as table 12-15 for TFR, using footnotes:

- Only adverse events from TFR phase are included in this table. Specific groups are alphabetically presented; preferred terms are sorted within each group in descending frequency of 'All grades' column. Percentage based on population number (N). Treatment Arm 1/Arm 2: 24/36 months, Re-treatment max Arm 1/Arm 2: 36/24 months. A patient with multiple occurrences of an AE is counted only once in the AE category. A patient with multiple AE within a primary system organ class is counted only once in the total row. AE of special interest CVEs (IHD), CVEs (PAOD), CVEs (ICD) and CVEs (others) are based on grouped MedDRA terms as described in the Case Retrieval Sheet.

Source: Post-text table: 14.3.1-6.7.1

# Table 12-17 Treatment-emergent adverse events incidence leading to study drug discontinuation by system organ class and preferred term during pre-randomization Induction/Consolidation phase – overall and maximum grade 3/4 –Full Analysis Set


CAMN107AIC05

| | Arı | m 1 | | | To | tal |
|---|---|---|---|---|---|---|
| | N= | XXX | N=x | XX | N= | XXX |
| Primary system organ | All | Grade | All | Grade | All | Grade |
| class | grades | 3/4 | grades | 3/4 | grades | 3/4 |
| Preferred term | n (%) | n (%) | n (%) | n (응) | n (%) | n (%) |
| Any Primary system organ class | xx (xx.x) | xx (xx.x) | | | xx (xx.x) | xx (xx.x) |
| Cardiac disorders | xx (xx.x) | xx (xx.x) | | | xx (xx.x) | xx (xx.x) |
| Angina pectoris | xx (xx.x) | xx (xx.x) | | | xx (xx.x) | xx (xx.x) |
| Bradycardia NOS | xx (xx.x) | xx (xx.x) | | | xx (xx.x) | xx (xx.x) |
| Oedema NOS | xx (xx.x) | xx (xx.x) | | | xx (xx.x) | xx (xx.x) |
| Tachycardia NOS | xx (xx.x) | xx (xx.x) | | | xx (xx.x) | xx (xx.x) |

- For patient # \_\_\_\_\_, due to reconciliation discrepancies, safety database reported AE term "Endometriosis" as a SAE, while in clinical database this AE was not recorded as an SAE.

<sup>-</sup> Only TEAEs from pre-rand. ind./cons. phase have been included. Prim. SOC are presented alphab.; PTs are sorted within prim. SOC in descending freq. of 'All grades' column. Perc. based pop. number (N). Treatment Arm 1/Arm 2: 24/36 months, Re-trt max Arm 1/Arm 2: 36/24 months. A patient with mult. occur. of an AE is counted only once in the AE category. A patient with mult. AEs within a primary SOC is counted only once in the total row. AEs occurring more than 30 days after last study trt. exp. date are not summarized. Pat. # reported as disc. Ind/Cons phase due to AE "Blast Crisis"- G2, should have been reported as disc. Ind/Cons phase due to Disease Progression, progression to Blast Crisis, as per Prot. Source: Post-text table: 14.3.1-5.1.1

Table 12-18 Treatment-emergent adverse events incidence leading to study drug discontinuation by system organ class and preferred term during post-randomizationphase (ARM 2) – overall and maximum grade 3/4 – Subset of Full Analysis Set randomized to Arm 2

| | Ar | m2 |
|--------------------------------|-----------|-----------|
| | N=> | XXX |
| Primary system organ class | All | Grade |
| Preferred term | grades | 3/4 |
| | n (응) | n (응) |
| Any Primary system organ class | xx (xx.x) | xx (xx.x) |
| Cardiac disorders | xx (xx.x) | xx (xx.x) |
| Angina pectoris | xx (xx.x) | xx (xx.x) |
| Bradycardia NOS | xx (xx.x) | xx (xx.x) |
| Oedema NOS | xx (xx.x) | xx (xx.x) |
| Tachycardia NOS | xx (xx.x) | xx (xx.x) |
| • • • | | |

<sup>-</sup> Only TEAEs from post-rand. Cons. phase (ARM 2) are included in this table. Primary system organ classes are presented alphabetically; preferred terms are sorted within primary system organ class in descending frequency of 'All grades' column. Percentage based on the number of patients included in the analysis population (N). Treatment post-randomization Arm 2: 12 months, treatment free remission max Arm 2: 24 months. A patient with multiple occurrences counted only once in the AE category. A patient with multiple AEs within a primary system organ class is counted only once in the total row. AEs occurring more than 30 days after last study treatment exposure date are not summarized.

Source: Post-text table: 14.3.1-5.2.1

Table 12-19 On treatment deaths, by system organ class and preferred term during pre-randomization Induction/Consolidation phase - Safety Set

| Primary system organ class<br>Principal cause of death | Arm 1<br>N=xxx<br>n (%) | N=xxx<br>n (%) | Total<br>N=xxx<br>n (%) |
|---|---|---|---|
| Any Primary system organ class | xx (xx.x) | | xx (xx.x) |
| Primary system organ class 1 | xx (xx.x) | | xx (xx.x) |
| Preferred term 1 | xx (xx.x) | | xx (xx.x) |
| Preferred term 2 | xx (xx.x) | • • • | xx (xx.x) |

Primary system organ classes are alphabetically presented; preferred terms are sorted within primary system organ class in descending frequency.

Source: Post-text table: 14.3.1-9.1

<sup>-</sup> Percentage based on the number of patients included in the analysis population (N).

<sup>-</sup> Treatment Arm 1/Arm 2: 24/36 months, Re-treatment max Arm 1/Arm 2: 36/24 months.

<sup>-</sup> Deaths up to 30 days after last study treatment exposure date are all included

- For patient date of death was imputed to "for the purpose of this table only."

"" for the purpose of this table only."

# Table 12-20 On treatment deaths, by system organ class and preferred term during post-randomization consolidation phase (ARM 2) – Subset of Safety Set randomized to Arm 2

| Primary system organ class<br>Principal cause of death | Arm 2<br>N=xxx<br>n (%) |
|---|---|
| Any Primary system organ class | xx (xx.x) |
| Primary system organ class 1 | xx (xx.x) |
| Preferred term 1 | xx (xx.x) |
| Preferred term 2 | xx (xx.x) |
| • • • | |

<sup>-</sup> Primary system organ classes are alphabetically presented; preferred terms are sorted within primary system organ class in descending frequency.

- Percentage based on the number of patients included in the analysis population (N).
- Treatment post-randomization Arm 2: 12 months, Re-treatment max Arm 2: 24 months.
- Deaths up to 30 days after last study treatment exposure date are all included. Source: Post-text table: 14.3.1-9.2

# Table 12-21 On treatment deaths, by system organ class and preferred term during re-treatment phase – Subset of Safety Set entering the re-treatment phase

<< Programming note: Same shell as table 10-15.1.1 presenting only Arm 1, Arm 2 and Total for Re-treatment>>

Primary system organ classes are alphabetically presented; preferred terms are sorted within primary system organ class in descending frequency.

- Only deaths occurring during the treatment period (between the first day of study drug intake and up to 30 days after last study drug intake) are presented.
- Percentage based on the number of patients included in the analysis population (N).
- Treatment Arm 1/Arm 2: 24/36 months, Re-treatment max Arm 1/Arm 2: 36/24 months. Source: Post-text table: 14.3.1-9.3

### Listing 12-1 Listing of deaths - Full Analysis Set

| Country/<br>Center/<br>Patient/<br>Arm | Age/<br>Sex/<br>Race | Date<br>of<br>last<br>dose | Study<br>day of<br>last<br>dose | Date of<br>death<br>(phase) | Study day<br>of death | Number<br>days<br>since<br>last dose | Principal<br>cause of death<br>reported/<br>Preferred term |
|---|---|---|---|---|---|---|---|
| XXX/0XXX<br>/0XXXX/X | XX/X<br>/XX | DDMMM<br>YYYY | XX | DDMMMYYYY<br>(IND/CONS1/C<br>ONS2/TFR/<br>RE-TRT) | xx | xx | XXXXXXXXX/XXX<br>XXXX |
| XXX/0XXX<br>/0XXXX/X | XX/X<br>/XX | DDMMM<br>YYYY | XX | DDMMMYYYY<br>(IND/CONS1/C<br>ONS2/TFR/<br>RE-TRT) | xx # | xx * | XXXXXXXXX/XXX<br>XXXX |

<sup>-</sup> Arm: 1: Arm 1; 2: Arm 2; 3: Not Randomized. Phase: IND = ind. phase (0-12 m), CONS1 = pre-rand. cons. phase (12-24 m), CONS2 = post-rand. cons. phase (ARM 2)(24-36 m), TFR=treat. free remission phase and RE-TRT=re-treat. phase. Phase displayed indicates in which end of phase page the death has been recorded as the primary reason to discontinue the study. If missing then death has been recorded in survival follow-up CRF pages. Study day relative to the first day of treatment (day 1).\*event occurred more than 30 days after last study treatment exposure date. # Death occurring outside the treatment emergent period - Number of days since last dose = day of death - day of last dose + 1.

<sup>-</sup> Number of days since last dose = day of death - day of last dose + 1 Source: Post-text listing: 14.3.2-1.1

Figure 11-1 Primary endpoint, Bar plot MR4.0 at 12 months of TFR phase
-Subset of Full Analysis Set entering the TFR phase



Source: Post-text figure: 14.2-16

Programming Note: Use black color but different patterns for each bar.

Figure 11-2 Kaplan-Meier analysis of treatment-free survival during the TFR phase –Subset of Full Analysis Set entering the TFR phase



#### Programming note:

The axis label should "Time since start of TFR phase (months)" Months 24-60 for Arm 1, Months 36-60 for Arm 2

Vertical (Y-Axis) label "Prop. of pts. without treatment" Source: Post-text figure: 14.2-17.2

## 3.2 Shells and specifications for Sections 14 and 16 of the CSR

Section 14 – tables, figures and graphs referred to but not included in the text


CAMN107AIC05

Section 14.1 - Demographic data

Figures (Section 14.1)

Not applicable

Tables (Section 14.1)

Table 14.1-1.1 Enrollment by country and center - All patients

| Country | Arm 1 | Arm 2 | Randomized | Not Randomized N=xx | Not | Total |
|---|---|---|---|---|---|---|
| Center | N=xx | N=xx | N=xx | | treated | N=xx |
| All countries | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Denmark (2) xxxx xxxxx | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx (xx.x) | xx(xx.x) |
| | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx (xx.x) | xx(xx.x) |
| France (8) xxxx xxxxx | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx (xx.x) | xx (xx.x) | xx(xx.x) |
| | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx (xx.x) | xx (xx.x) | xx(xx.x) |

<sup>-</sup> Arm 1: ARM 1: the nilotinib 24 months treatment arm.

The numbers in parentheses provide the number of centers for the country.

#### << Programming note:

The number of centers per country will always be indicated in parenthesis. Percentages are calculated out of the all screened patients>>

<sup>-</sup> Arm 2: ARM 2: the nilotinib 36 months treatment arm.

<sup>-</sup> Randomized: Arm 1+ Arm 2.

<sup>-</sup> Not Randomized: Screened and treated but Not Randomized patients.

<sup>-</sup> Not Treated: Screen Failures.

#### Table 14.1-1.2 Randomization by country and center – Randomized patients

| Country<br>Center | Arm 1<br>N=xx | Arm 2<br>N=xx | Total<br>N=xx |
|---|---|---|---|
| All countries | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Denmark (2)<br>xxxx<br>xxxx | , , | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) |
| France (8) xxxx xxxx | , , | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) |
| Etc | | | |

<sup>-</sup> Arm 1: ARM 1: the nilotinib 24 months treatment arm.

<sup>-</sup> Arm 2: ARM 2: the nilotinib 36 months treatment arm.

<sup>-</sup> Randomized: Arm 1+ Arm 2.

<sup>-</sup> The numbers in parentheses provide the number of centers for the country.

<sup>-</sup> Percentage is based on N.

<sup>-</sup> Patients randomized to Arm 1 have 24 months of treatment and a maximum of 36 months of re-treatment.

<sup>-</sup> Patients randomized to Arm 2 have 36 months of treatment and a maximum of 24 months of re-treatment.

<sup>&</sup>lt;< Programming note: The number of centers per country will always be indicated in parenthesis. Percentages are calculated out of the FAS patients>>

# Table 14.1-1.3 Patient disposition (Screening failures), All patients

| Disposition Reason | Total<br>N=XXX |
|--------------------------------------|----------------|
| Screened patients | XXX (100.0) |
| Screened successfully | ZZZ |
| Re-screened | YYY |
| Screen Failures | FFF |
| Reason for Screen failure | |
| As per protocol | XX |
| Scheduling conflict | XX |
| Other | XX |
| Inclusion/Exclusion criteria not met | XX |
| Inclusion Criteria* | |
| XXXXXXXXX | XX |
| XXXXXXXXX | XX |
| ••• | |
| XXXXXXXXX | XX |
| Exclusion Criteria* | |
| xxxxxxxxx | XX |
| xxxxxxxxx | xx |
| xxxxxxxxx | xx |

<sup>\*</sup> Patients enrolled but excluded due to Inclusion/Exclusion Criteria. Multiple reasons for screen failure for patients.

Novartis Confidential Page 142 RAP Module 7.1 Confidential Protocol No CAMN107AIC0

#### Programing Note:

Present only specific Incl/Excl criteria text, do not use numbers since ICX may correspond to different text depending on Protocol version.

Present Reason for Screen failure Reason for patients enrolled but excluded due to Inclusion/Exclusion Criteria. Use intents before labels of subcategories as in the shell.

Table 14.1-2.1 Patient disposition during Induction/Consolidation phase and post-Randomization Consolidation phase -Enrolled patients

| Disposition<br>Reason | | arm 1<br>N=xx | | Arm 2<br>N=xx | | domized<br>N=xx | | andomized<br>N=xx | | Total<br>N=xx |
|---|---|---|---|---|---|---|---|---|---|---|
| Patients enrolled | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | xx | (xx.x) | XX | (xx.x) |
| Patients not-treated[1] | | | | | | | | | | |
| Primary reason for study discontinuation | | | | | | | | | | |
| Adverse event(s) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) |
| Abnormal laboratory value(s) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) |
| Abnormal test procedure result(s) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) |
| Pregnancy | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) |
| Protocol deviation | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) |
| Subject withdrew consent | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) |
| Lost to follow-up | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) |
| Administrative problems | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) |
| Disease progression (CML) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) |
| Unstable MR4.0 | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) |
| New cancer (CML) therapy | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) |
| Relapse loss MMR/MR4 | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) |
| Other | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | | |
| Death | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) |
| Patients treated [2] | | | | | | | | | | |
| Patients treated | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) |
| Discontinued from treatment | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) |
| Primary reason for study discontinuation | | | | | | | | | | |
| Adverse event(s) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) |
| Abnormal laboratory value(s) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) |

<sup>-</sup> Percentage is based on N

<sup>[1]</sup> Patients who discontinued study after enrollment without taking study drug.

<sup>[2]</sup> Patients who discontinued study during Induction/Consolidation phase.

<sup>- 15</sup> patients from ARM 2 discontinued during post-Randomization Consolidation phase.

<sup>-</sup> Patient # randomized to Arm 1 at and discontinued Ind/cons at the same day for '

<sup>-</sup> Patient # reported as disc. Ind/Cons phase due to AE "Blast Crisis"- G2, should have been reported as disc. Ind/Cons phase due to Disease Progression, progression to Blast Crisis, as per Prot.

#### Table 14.1-2.2 Patient disposition in each randomized arm – Full Analysis Set

Page 1 on 2

| Disposition | N= | xx |
|---|---|---|
| | n | (%) |
| Number of patients with no major deviation to protocol | XX | (xx.x) |
| Randomized patients | XX | (xx.x) |
| Arm 1 Nilotinib 24-month treatment arm [1] | XX | (xx.x) |
| Patients completed the consolidation phase [2] | XX | (xx.x) |
| Patients discontinued before TFR phase [2] | XX | (xx.x) |
| Patients entered in the TFR phase [2] | XX | (xx.x) |
| Patients who completed the TFR phase (36 months) [3] | XX | (xx.x) |
| Patients in the TFR phase with 6 months (i.e. 213 days) without relapse [3] | XX | (xx.x) |
| Patients in the TFR phase with 12 months (i.e. 411 days) without relapse [3] | XX | (xx.x) |
| Patients discontinued TFR phase without entering re-treatment phase [3] | XX | (xx.x) |
| - entering in survival follow-up period [4] | XX | (xx.x) |
| - completing the survival follow-up and the 5 years study period [4] | XX | (xx.x) |
| - completing the survival follow-up before the 5 years study period [4] | XX | (xx.x) |
| <ul> <li>discontinued from the study without survival follow-up [4]</li> </ul> | XX | (xx.x) |
| Patients discontinued TFR and entered in the re-treatment phase [3] | XX | (xx.x) |
| Patients discontinued the re-treatment phase [5] | XX | (xx.x) |
| - completing the survival follow-up and the 5 years study period [6] | XX | (xx.x) |
| - completing the survival follow-up before the 5 years study period [6] | XX | (xx.x) |
| - discontinued from the study without survival follow-up [6] | XX | (xx.x) |
| Patients who completed the re-treatment phase [5] | XX | (xx.x) |

<sup>[1]</sup> Percentage based on the number of patients included in the analysis population (N).

Patient # remained in TFR until EoS. EOP TFR was erroneously completed and data not reconciled.

<sup>[2]</sup> Percentage based on the number of patients randomized at each treatment arm.

<sup>[3]</sup> Percentage based on the number of patients entered in the TFR phase at each treatment arm.

<sup>[4]</sup> Percentage based on the number of patients discontinued TFR phase without entering in the re-treatment phase.

<sup>[5]</sup> Percentage based on the number of patients entered in the re-treatment phase.

<sup>[6]</sup> Percentage based on the number of patients discontinued the re-treatment phase.

Protocol deviation excluding patient from per protocol analysis set is defined as major protocol deviation (PD severity codes: 0, 1, 5, 8).

Page 2 on 2

| isposition | N=xx<br>n (%) |
|---|---|
| Arm 2 Nilotinib 36-month treatment arm [1] | xx (xx.x) |
| Patients completed the consolidation phase [2] | xx (xx.x) |
| Patients entered in the TFR phase [2] | xx (xx.x) |
| Patients discontinued before TFR phase [2] | xx (xx.x) |
| Patients who completed the TFR phase (24 months) [3] | xx (xx.x) |
| Patients in the TFR phase with 6 months (i.e. 213 days) without relapse [3] | xx (xx.x) |
| Patients in the TFR phase with 12 months (i.e. 411 days) without relapse [3] | xx (xx.x) |
| Patients discontinued TFR phase without entering re-treatment phase [3] | xx (xx.x) |
| - entering in survival follow-up period [4] | xx (xx.x) |
| - completing the survival follow-up and the 5 years study period [4] | xx (xx.x) |
| - completing the survival follow-up before the 5 years study period [4] | xx (xx.x) |
| - discontinued from the study without survival follow-up [4] | xx (xx.x) |
| Patients discontinued TFR and entered in the re-treatment phase [3] | xx (xx.x) |
| Patients discontinued the re-treatment phase [5] | xx (xx.x) |
| - completing the survival follow-up and the 5 years study period [6] | xx (xx.x) |
| - completing the survival follow-up before the 5 years study period [6] | xx (xx.x) |
| - discontinued from the study without survival follow-up [6] | xx (xx.x) |
| Patients who completed the re-treatment phase [5] | xx (xx.x) |

- [1] Percentage based on the number of patients included in the analysis population (N).
- [2] Percentage based on the number of patients randomized at each treatment arm.
- [3] Percentage based on the number of patients entered in the TFR phase at each treatment arm.
- [4] Percentage based on the number of patients discontinued TFR phase without entering in the re-treatment phase.
- [5] Percentage based on the number of patients entered in the re-treatment phase.
- [6] Percentage based on the number of patients discontinued the re-treatment phase.

Protocol deviation excluding patient from per protocol analysis set is defined as major protocol deviation (PD severity codes: 0, 1, 5, 8).

Patient # rem

remained in TFR until EoS. EOP TFR was erroneously completed and data not reconciled.

#### << Programming note:

Enrolled patients (who signed IFC and who met IE criteria): present in IFC dataset (with IFC1D not missing) and IECELI1C=yes in IEC dataset

Treated patients: at least one piece of data in DAR

Randomized patients: IECELIC1 (Subject eligible for randomization?)=yes in CRI dataset

Arm 1: RND1C=1 in IVRS dataset

Arm 1 who completed the TFR phase: RND1C=1 in IVRS dataset, and remaining in TFR up to EOS (ie in CMP, subject has VISNAM1A= V403-EOS and SBJCMP1C (Subject completed 5 years study period?)=yes)

Arm 1 who entered the re-treatment phase: RND1C=1 in IVRS dataset, and in CMP, Patient should have taken drug in RT phase.Arm 2: RND1C=2 in IVRS dataset

Arm 2 eligible for TFR: RND1C=2 in IVRS dataset, and IECELIC2 (Subject eligible for TFR phas?)=yes in CRI dataset

Arm 2 who completed the TFR phase: RND1C=2 in IVRS dataset, and remaining in TFR up to EOS (ie in CMP, subject has VISNAM1A= V403-EOS and SBJCMP1C (Subject completed 5 years study period?)=yes)

Arm 2 who entered the re-treatment phase: RND1C=2 in IVRS dataset, Patient should have taken drug in RT phase.>>

# Table 14.1-2.2.1 Patient disposition – Enrolled patients in LSC substudy

| Disposition | N=xx<br>n (%) |
|---|---|
| Patients enrolled in the induction/consolidation phase | xx (xx.x) |
| Patients Not Randomized | xx (xx.x) |
| Patients who received at least one dose of nilotinib | xx (xx.x) |
| Randomized patients Nilotinib 24-month treatment arm (Arm 1) | xx (xx.x)<br>xx (xx.x) |
| Nilotinib 36-month treatment arm (Arm 2) | xx (xx.x) |
| Patients with no major deviation to protocol | xx (xx.x) |

<sup>-</sup> Percentage is based on N

<sup>-</sup> LSC: Leukemic Stem Cells. Enrolled in LSC are patients signed the LSC ICF.

## Table 14.1-2.3 Analysis sets -All patients

| | All patients<br>N=xx |
|----------------------------|----------------------|
| Analysis set | n (%) |
| Screened patients | xx (xx.x) |
| Screened succesfully | xx (xx.x) |
| Re-screened | xx (xx.x) |
| Screen failures | xx (xx.x) |
| Enrolled patients | xx (xx.x) |
| Randomized patients* | xx (xx.x) |
| Not Randomized patients | xx (xx.x) |
| Enrolled patients (FAS) * | xx (xx.x) |
| Randomized patients* | xx (xx.x) |
| Not Randomized patients* | xx (xx.x |
| Safety Set* | xx (xx.x) |
| Per Protocol Analysis Set* | xx (xx.x) |

<sup>-</sup> Randomized patients are all patients meeting eligibility criteria for randomization (i.e. achieved a sustained MR4.0 for at least 12 months in the Induction/Consolidation phase of the study).

<sup>-</sup> Full Analysis Set (FAS) comprises all subjects who are enrolled, excluding patients with PD severity codes: 0, 8.

<sup>-</sup> Safety Set consists of all patients who received at least one dose of study drug, excluding patients with PD severity codes: 0, 5, 8.

Per Protocol Analysis Set (PPS) comprises all subjects who are enrolled without major protocol deviation (PD severity codes: 0, 1, 5, 8)

<sup>\*</sup> Patients without major PD.

# Table 14.1-2.4 Not Randomized patients - Enrolled patients

| | | Cotal<br>(N=XX)<br>n (%) |
|---|---|---|
| Not Randomized Patients | | XX |
| Reasons | | |
| Patient with last assessment < MR4.0 | xx | (xx.x) |
| Patient with < 4 times MR4.0, out of 5 times MR4.0 | xx | (xx.x) |
| Patient with no MR4.0, out of 5 times MR4.0 | XX | (xx.x) |
| Patient with 1 time MR4.0, out of 5 times MR4.0 | | (xx.x) |
| Patient with 2 times MR4.0, out of 5 times MR4.0 | XX | (xx.x) |
| Patient with 3 times MR4.0, out of 5 times MR4.0 | XX | (xx.x) |
| Patient with < 4 times MR4.0, out of 5 times MR4.0 and last assessment < MR4.0 | xx | (xx.x) |
| Patient with no MR4.0, out of 5 times MR4.0 | XX | (xx.x) |
| Patient with 1 time MR4.0, out of 5 times MR4.0 | XX | (xx.x) |
| Patient with 2 times MR4.0, out of 5 times MR4.0 | XX | (xx.x) |
| Patient with 3 times MR4.0, out of 5 times MR4.0 | XX | (xx.x) |
| Patient with 4 times MR4.0, out of 5 times, MR4.0 but last assessment $<$ MR4.0 | xx | (xx.x) |
| Patient with $<$ 4 times MR4.0 out of 5 times MR4.0, with last assessment MR4.0 | xx | (xx.x) |
| Other reason* | XX | (xx.x) |

<sup>\*</sup> Other reason not related to Molecular response, including: AE, ICF withdrew, PD, lost to follow up, death, etc.

# Table 14.1-2.5 Patient disposition, Overall and by year-phase -Enrolled patients

| Disposition<br>Reason | Arm 1<br>N=xx | Arm 2<br>N=xx | Randomized<br>N=xx | Not Randomized N=xx | Total<br>N=xx |
|---|---|---|---|---|---|
| Total | | | | | |
| Patients enrolled | xx (xx.x | ) xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Patients not-treated[1] | | | | | |
| Primary reason for study discontinuation | | | | | |
| Adverse event(s) | xx (xx.x | ) xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Abnormal laboratory value(s) | xx (xx.x | $)$ $\times \times (\times \times \times)$ | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Abnormal test procedure result(s) | xx (xx.x | ) $xx (xx.x)$ | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Pregnancy | xx (xx.x | ) $xx (xx.x)$ | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Protocol deviation | xx (xx.x | ) $xx (xx.x)$ | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Subject withdrew consent | xx (xx.x | ) xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Lost to follow-up | xx (xx.x | ) $xx (xx.x)$ | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Administrative problems | xx (xx.x | ) $xx (xx.x)$ | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Disease progression (CML) | xx (xx.x | ) $xx (xx.x)$ | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Unstable MR4.0 | xx (xx.x | ) $xx (xx.x)$ | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| New cancer (CML) therapy | xx (xx.x | ) $xx (xx.x)$ | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Death | xx (xx.x | ) xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Patients treated [2] | | | | | |
| Patients treated | xx (xx.x | ) $xx (xx.x)$ | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Discontinued from treatment | xx (xx.x | ) xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Primary reason for study discontinuation | | | | | |
| Adverse event(s) | xx (xx.x | ) xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Death | xx (xx.x | ) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

#### Induction-Consolidation 1st year

Patients not-treated[3]

Primary reason for study discontinuation

| Novartis<br>RAP Module 7.1 | Confidential<br>6-May-2021 (14:35) | Protocol No | Page 151<br>CAMN107AIC0 |
|---|---|---|---|
| Adverse event(s) | xx (xx.x) xx (xx.x) > | xx (xx.x) | xx (xx.x) |
| <br>Death | xx (xx.x) > | | <br>xx (xx.x) |
| Deach | ** (****) ** (****) * | (X (XX.X) XX (XX.X) | xx (xx.x) |
| Patients treated [2] Patients treated | xx (xx.x) xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Discontinued from treatment | , | xx (xx.x) | xx (xx.x)<br>xx (xx.x) |
| Primary reason for study discontinuation | | | |
| Adverse event(s) | , | xx (xx.x) | xx (xx.x) |
| Death | xx (xx.x) xx (xx.x) | <br>xx (xx.x) | xx (xx.x) |
| Induction-Consolidation 2nd year (pre-<br>randomization consolidation) | | | |
| Patients treated [2] | | | |
| Patients treated Discontinued from treatment | | xx (xx.x) | xx (xx.x)<br>xx (xx.x) |
| | AA (AA.A) AA (AA.A) Z | \(\lambda \lambda \lam | AA (AA.A) |
| Primary reason for study discontinuation Adverse event(s) | () | () | ( |
| Adverse event(s) | xx (xx.x) xx (xx.x) x | xx (xx.x) | xx (xx.x) |
| Death | xx (xx.x) xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3rd year of treatment (post-randomization consolidation) | | | |
| Patients treated [2] | | | |
| Patients treated Discontinued from treatment | | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) |
| Primary reason for study discontinuation | XX (XX.X) Z | (X (XX.X) | XX (XX.X) |
| Adverse event(s) | , , | xx (xx.x) | xx (xx.x) |
| Death | xx (xx.x) | <br>xx (xx.x) | xx (xx.x) |
| TFR period | | | |
| Patients entered TFR | | xx (xx.x) | xx (xx.x) |
| TFR ongoing | xx (xx.x) xx (xx.x) | xx (xx.x) | xx (xx.x) |

| Novartis<br>RAP Module 7.1 | Confident<br>6-May-2021 ( | | | Page 152<br>Protocol No CAMN107AIC0 |
|---|---|---|---|---|
| Patients Completed TFR | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Discontinued from TFR | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Primary reason for study discontinuation Adverse event(s) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| <br>Death | <br>xx (xx.x) | <br>xx (xx.x) | <br>xx (xx.x) | <br>xx (xx.x) |
| Primary reason for study discontinuation | () | (, | (, | ( |
| Re-treatment period | | | | |
| Patients entered re-treatment period | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Patients not-treated (during re-treatment) [4] Primary reason for study discontinuation | | | | |
| Adverse event(s) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Death | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Patients treated (during re-treatment) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Re-Treatment ongoing # | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Re-treatment completed | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Discontinued from treatment | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Primary reason for study discontinuation | , , | | | |
| Adverse event(s) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Death | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Survival follow-up period | | | | |
| Patients entered survival follow-up period | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Patients followed during survival follow-up | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Survival follow-up ongoing | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Survival follow-up completed | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Discontinued from survival follow-up | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Primary reason for death | | | | |
| CML | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

<sup>#</sup> Patients with treatment ongoing in Re-treatment phase at the time of DBL ddmmmyyyy.

<sup>-</sup> Percentage is based on N.

<sup>[1]</sup> Patients who discontinued study after enrollment without taking study drug.
[2] Patients who discontinued study during Induction/Consolidation phase, having received study drug.

- [3] Patients who discontinued study after enrollment without taking study drug, during  $1^{\rm st}$  year of Induction-Consolidation
- [4] Patients who discontinued study after start of re-treatment without taking study drug.
- Patient # reported as disc. Ind/Cons phase due to AE "Blast Crisis"- G2, should have been reported as disc. Ind/Cons phase due to Disease Progression, progression to Blast Crisis, as per Prot. Patient # remained in TFR until EoS. EOP TFR was erroneously completed and data not reconciled.

#### << Programming note:

Sort reason for discontinuation by decreasing frequency >>

# Table 14.1-2.6 Patients discontinued and reason for discontinuation – Full Analysis Set

| Disposition<br>Reason | Arm 1<br>N=xx | Arm 2<br>N=xx | Randomized<br>N=xx | Not Randomized<br>N=xx | Total<br>N=xx |
|---|---|---|---|---|---|
| Patients discontinued at any time-point after Randomization | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Primary reason for discontinuation [1] | | | | | |
| Adverse event(s) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Abnormal laboratory value(s) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Abnormal test procedure result(s) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Pregnancy | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Protocol deviation | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Subject withdrew consent | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Lost to follow-up | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Administrative problems | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Disease progression (CML) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Relapse (Loss of MMR/confirmed loss of MR4.0) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| New cancer (CML) therapy | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Death | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Patients discontinued before TFR [2] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Primary reason for discontinuation | | | | | |
| Adverse event(s) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Abnormal laboratory value(s) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Abnormal test procedure result(s) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Pregnancy | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Protocol deviation | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Subject withdrew consent | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Lost to follow-up | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Administrative problems | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Disease progression (CML) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Relapse (Loss of MMR/confirmed loss of MR4.0) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| New cancer (CML) therapy | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Death | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx (xx.x) | xx (xx.x) | xx (xx.x) | | xx (xx.x) |

| Planathia | 7 1 | 7 | Dan dan i a a | Mat Dandania ad | m - + - 1 |
|---|---|---|---|---|---|
| Disposition<br>Reason | Arm 1<br>N=xx | Arm 2<br>N=xx | Randomized<br>N=xx | Not Randomized<br>N=xx | Total<br>N=xx |
| | | | | IV-XX | |
| Patients entered in the TFR phase | xx (xx.x) | xx (xx.x) | xx (xx.x) | | xx (xx.x) |
| Patients discontinued from the TFR phase | xx (xx.x) | xx (xx.x) | xx (xx.x) | | xx (xx.x) |
| Primary reason for TFR discontinuation | | | | | |
| Adverse event(s) | xx (xx.x) | xx (xx.x) | xx (xx.x) | | xx (xx.x) |
| Abnormal laboratory value(s) | xx (xx.x) | xx (xx.x) | xx (xx.x) | | xx (xx.x) |
| Abnormal test procedure result(s) | xx (xx.x) | xx (xx.x) | xx (xx.x) | | xx (xx.x) |
| Pregnancy | xx (xx.x) | xx (xx.x) | xx (xx.x) | | xx (xx.x) |
| Protocol deviation | xx (xx.x) | xx (xx.x) | xx (xx.x) | | xx (xx.x) |
| Subject withdrew consent | xx (xx.x) | xx (xx.x) | xx (xx.x) | | xx (xx.x) |
| Lost to follow-up | xx (xx.x) | xx (xx.x) | xx (xx.x) | | xx (xx.x) |
| Administrative problems | xx (xx.x) | xx (xx.x) | xx (xx.x) | | xx (xx.x) |
| Disease progression (CML) | xx (xx.x) | xx (xx.x) | xx (xx.x) | | xx (xx.x) |
| Relapse (Loss of MMR/confirmed loss of MR4.0) | xx (xx.x) | xx (xx.x) | xx (xx.x) | | xx (xx.x) |
| New cancer (CML) therapy | xx (xx.x) | xx (xx.x) | xx (xx.x) | | xx (xx.x) |
| Death | xx (xx.x) | xx (xx.x) | xx (xx.x) | | xx (xx.x) |
| Other | xx (xx.x) | xx (xx.x) | xx (xx.x) | | xx (xx.x) |
| Patients entered in the re-treatment phase | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Patients discontinued from the re-treatment phase | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Primary reason for re-treatment discontinuation | | | | | |
| Adverse event(s) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Abnormal laboratory value(s) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Abnormal test procedure result(s) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Pregnancy | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Protocol deviation | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Subject withdrew consent | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Lost to follow-up | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Administrative problems | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Disease progression (CML) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| New cancer (CML) therapy | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Death | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Patients entered in the survival follow up | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

- Percentage based on the number of patients included in the analysis population (N).
- [1] Primary discontinuation reasons summarized are relative to each phase and thus one patient can have several reasons of discontinuation corresponding to discontinuations from different phases.
- [2] For treatment Arm 1 patients discontinued before TFR, may occur between Randomization and treatment administration.
- Patient # reported as disc. Ind/Cons phase due to AE "Blast Crisis"- G2, should have been reported as disc. Ind/Cons phase due to Disease Progression, progression to Blast Crisis, as per Prot. Patient # remained in TFR until EoS. EOP TFR was erroneously completed and data not reconciled.

#### << Programming note:

Patients entered in TFR phase: corresponds to Arm 1 patients randomized (RND1C=1 in IVRS dataset) + Arm 2 patients eligible for TFR phase (RND1C=2 in IVRS dataset, and IECELIC2 (Subject eligible for TFR phase?)=yes in CRI dataset)

Patients discontinued from TFR phase: in CMP, subject has VISNAM1A= V401-EOP-TFR + DCNRSN1C for reason for discontinuation from TFR phase

Patients entered in re-treatment phase: in CMP, subject has VISNAM1A=V401-EOP-TFR and RTMTPH1C (Does the subject enter the retreatment phase?)=yes

Patients discontinued from re-treatment phase: in CMP, subject has VISNAM1A= V402-EOP-RT + DCNRSN1C for reason for discontinuation from re-treatment phase.

Sort reasons for discontinuation by descending frequency.>>

#### Table 14.1-2.6.1 Patients discontinued and reason for discontinuation, SDV sensitivity – Full Analysis Set

<< Programming note: Same shell as table 14.1-2.6, for SDV sensitivity analysis>>

- Percentage based on the number of patients included in the analysis population (N).
- [1] Primary discontinuation reasons summarized are relative to each phase and thus one patient can have several reasons of discontinuation corresponding to discontinuations from different phases.
- [2] For treatment Arm 1 patients discontinued before TFR, may occur between Randomization and treatment administration.
- SDV sensitivity: Excluding patient visits involved in SDV issues during final data review due to COVID-19.
- Patient # reported as disc. Ind/Cons phase due to AE "Blast Crisis"- G2, should have been reported as disc. Ind/Cons phase due to Disease Progression, progression to Blast Crisis, as per Prot. Patient # remained in TFR until EoS. EOP TFR was erroneously completed and data not reconciled.

Table 14.1-2.7 Summary of TFR phase – Full Analysis Set

| TFR | Arm 1<br>N=xx | Arm 2<br>N=xx | Total<br>N=xx |
|---|---|---|---|
| Number of patients entering the TFR phase | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of patients in TFR phase at Month 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of patients in TFR phase at Month 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of patients in TFR phase at Month 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of patients in TFR phase at Month 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of patients in TFR phase at Month 5 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of patients in TFR phase at Month 6 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of patients in TFR phase at Month 8 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of patients in TFR phase at Month 10 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of patients in TFR phase at Month 12 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of patients in TFR phase at Month 15 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of patients in TFR phase at Month 18 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of patients in TFR phase at Month 21 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of patients in TFR phase at Month 24 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of patients in TFR phase at Month 27 | xx (xx.x) | | xx (xx.x) |
| Number of patients in TFR phase at Month 30 | xx (xx.x) | | xx (xx.x) |

|----------------|--------------------|-------------------------|
| RAP Module 7.1 | 6-May-2021 (14:35) | Protocol No CAMN107AIC0 |

| Number | of | patients | in | TFR | phase | at | Month | 33 | XX | (xx.x) | XX | (xx.x) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Number | of | patients | in | TFR | phase | at | Month | 36 | XX | (xx.x) | XX | (xx.x) |

- Percentage based on the number of patients included in the analysis population (N).
- Patients randomized to Arm 1 have a maximum of 36 months of TFR phase.
- Patients randomized to Arm 2 have a maximum of 24 months of TFR phase.
- Month corresponds to time-window as defined in the RAP Module 3.

#### Table 14.1-2.7.1 Summary of TFR phase, SDV sensitivity – Full Analysis Set

<< Programming note: Same shell as table 14.1-2.7, for SDV sensitivity analysis>>

#### Add footnote:

- SDV sensitivity: Excluding patient visits involved in SDV issues during final data review due to COVID-19.

Table 14.1-2.8 Summary of re-treatment phase – Full Analysis Set

| Re-treatment | Arm 1<br>N=xx | Arm 2<br>N=xx | Total<br>N=xx |
|---|---|---|---|
| Number of Full Analysis Set entering the re-treatment phase | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of patients in re-treatment phase at Week 6 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of patients in re-treatment phase at Month 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of patients in re-treatment phase at Month 6 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of patients in re-treatment phase at Month 9 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of patients in re-treatment phase at Month 12 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of patients in re-treatment phase at Month 15 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of patients in re-treatment phase at Month 18 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of patients in re-treatment phase at Month 21 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of patients in re-treatment phase at Month 24 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of patients in re-treatment phase at Month 27 | xx (xx.x) | | xx (xx.x) |
| Number of patients in re-treatment phase at Month 30 | xx (xx.x) | | xx (xx.x) |
| Number of patients in re-treatment phase at Month 33 | xx (xx.x) | | xx (xx.x) |
| Number of patients in re-treatment phase at Month 36 | xx (xx.x) | | xx (xx.x) |

<sup>-</sup> Percentage based on the number of patients included in the analysis population (N).

<sup>-</sup> Patients randomized to Arm 1 have a maximum of 36 months of TFR phase.

<sup>-</sup> Patients randomized to Arm 2 have a maximum of 24 months of re-treatment phase.

<sup>-</sup> Week or Month corresponds to time-window as defined in the RAP Module 3.

### Table 14.1-2.8.1 Summary of re-treatment phase, SDV sensitivity – Full Analysis Set

<< Programming note: Same shell as table 14.1-2.8, for SDV sensitivity analysis>>

#### Add footnote:

- SDV sensitivity: Excluding patient visits involved in SDV issues during final data review due to COVID-19.

Table 14.1-2.9 Summary of patients with relapse during the TFR phase but no entering re-treatment phase — Subset of Full Analysis Set entering the TFR phase

| Relapse | Arm 1<br>N=xx | Arm 2<br>N=xx | Total<br>N=xx |
|---|---|---|---|
| Number of patients relapse but not enter the re-treatment phase | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of patients relapse but not enter re-treatment phase at Week 6 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of patients relapse but not enter re-treatment phase at Month 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of patients relapse but not enter re-treatment phase at Month 6 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of patients relapse but not enter re-treatment phase at Month 9 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of patients relapse but not enter re-treatment phase at Month 12 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of patients relapse but not enter re-treatment phase at Month 15 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of patients relapse but not enter re-treatment phase at Month 18 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of patients relapse but not enter re-treatment phase at Month 21 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of patients relapse but not enter re-treatment phase at Month 24 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of patients relapse but not enter re-treatment phase at Month 27 | xx (xx.x) | | xx (xx.x) |
| Number of patients relapse but not enter re-treatment phase at Month 30 | xx (xx.x) | | xx (xx.x) |
| Number of patients relapse but not enter re-treatment phase at Month 33 | xx (xx.x) | | xx (xx.x) |
| Number of patients relapse but not enter re-treatment phase at Month 36 | xx (xx.x) | | xx (xx.x) |
| Number of patients relapse but not enter the re-treatment phase immediately, but entered at re-treatment at a later stage. | xx (xx.x) | xx (xx.x) | xx (xx.x) |

NovartisConfidentialPage 162RAP Module 7.16-May-2021 (14:35)Protocol No CAMN107AIC0

- Percentage based on the number of patients included in the analysis population (N).
- Patients randomized to Arm 2 have a maximum of 24 months of re-treatment phase.
- Week or Month corresponds to time-window as defined in the RAP Module 3.
- Classification to each specific time window was based on time between Relapse and Re-treatment for patients with Re-treatment and time between Relapse and Last contact date, for patients with no Re-treatment at all.
- Due to the fact that only standard time points presented, any events occurred outside those standard time windows, although counted in "relapse but not enter the re-treatment phase" total category, were not presented in the following categories.

Table 14.1-3.1 Demographic and characteristics at baseline– Full Analysis Set

| Characteristics at baseline | Arm 1<br>N=xx | Arm 2<br>N=xx | Randomized<br>N=xx | Not Randomized<br>N=xx | Total<br>N=xx | Comparison\$<br>p-value# |
|---|---|---|---|---|---|---|
| Age at baseline visit(Years) - n (%) < 65 >= 65 Missing | xx (xx.x)<br>xx (xx.x)<br>xx | xx (xx.x)<br>xx (xx.x)<br>xx | xx (xx.x)<br>xx (xx.x)<br>xx | xx (xx.x)<br>xx (xx.x)<br>xx | xx (xx.x)<br>xx (xx.x)<br>xx | 0.xxx |
| Age at baseline visit (Years) | | | | | | |
| n | XXX | XXX | XXX | XXX | XXX | 0.xxx |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| SD | X.XX | X.XX | X.XX | X.XX | X.XX | |
| 25th Percentile | XX.X | XX.X | XX.X | XX.X | XX.X | |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | |
| 75th Percentile | XX.X | XX.X | XX.X | XX.X | XX.X | |
| Min-Max | xx-xx | XX-XX | XX-XX | XX-XX | XX-XX | |
| Gender - n (%) Female Male Missing | xx (xx.x)<br>xx (xx.x)<br>xx | xx (xx.x)<br>xx (xx.x)<br>xx | xx (xx.x)<br>xx (xx.x)<br>xx | xx (xx.x)<br>xx (xx.x)<br>xx | xx (xx.x)<br>xx (xx.x)<br>xx | 0.xxx* |
| If female, child bearing potential - n (%) | | | | | | |
| Able to bear children | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | 0.xxx |
| Premenarche | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | 0 • NNN |
| Post menopausal | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Sterile - of child bearing age | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Missing | XX (XX:X) | XX (XX:X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | |
| Race - n (%) | | | | | | |
| Caucasian | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | 0.xxx |
| Black | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Asian | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Native American | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| North African descent | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Unknown | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Other | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Missing | XX | XX | XX | XX | XX | |

| Characteristics at baseline | Arm 1 | Arm 2 | Randomized | Not Randomized | Total | Comparison\$ |
|---|---|---|---|---|---|---|
| | N=xx | N=xx | N=xx | N=xx | N=xx | p-value# |
| <b>-</b> 1 | | | | | | |
| Body mass index (kg/m2) - n (%) | , | , | , | , | , | 0 |
| Very severely underweight | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | 0.xxx |
| Severely underweight | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Underweight | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Normal | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Overweight | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Obese class I | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Obese class II | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Obese class III | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Missing | XX | XX | XX | XX | XX | |
| Body mass index (kg/m2) | | | | | | |
| n | XXX | XXX | XXX | XXX | XXX | 0.xxx |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| SD | X.XX | X.XX | X.XX | x.xx | X.XX | |
| 25th Percentile | XX.X | XX.X | XX.X | XX.X | XX.X | |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | |
| 75th Percentile | XX.X | XX.X | XX.X | XX.X | XX.X | |
| Min-Max | xx-xx | xx-xx | xx-xx | xx-xx | xx-xx | |
| F000 | | | | | | |
| ECOG performance Status (WHO) - n (%) | | | | | | |
| 0 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | 0.xxx |
| 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Missing | XX | XX | XX | XX | XX | |
| Family history - n (%) | | | | | | |
| Diabetes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Hypertension | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Dyslipidemia | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x) | |
| Cardiac events | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | |
| Cerebrovascular events | | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | , , | xx (xx.x)<br>xx (xx.x) | |
| Peripheral arterial disease | 1 1 | | | xx (xx.x) | , , | |
| - | , , | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Missing | XX | XX | XX | XX | XX | |

| Characteristics at baseline | Arm 1<br>N=xx | Arm 2<br>N=xx | Randomized<br>N=xx | Not Randomized<br>N=xx | Total<br>N=xx | Comparison\$<br>p-value# |
|---|---|---|---|---|---|---|
| Smoking history - n (%) | | | | | | |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | 0.xxx |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Ex-smoker | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Missing | xx | xx | XX | XX | XX | |
| If ex-smoker, time since stopped smoking | | | | | | |
| (months) | XXX | XXX | XXX | XXX | XXX | 0.xxx |
| n | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Mean | X.XX | X.XX | X.XX | X.XX | X.XX | |
| SD | XX.X | XX.X | XX.X | XX.X | XX.X | |
| 25th Percentile | XX.X | XX.X | XX.X | XX.X | XX.X | |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | |
| 75th Percentile | XX-XX | XX-XX | XX-XX | XX-XX | XX-XX | |
| Min-Max | | | | | | |
| If smoker or ex-smoker, use of tobacco | | | | | | |
| product in the past month - n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | 0.xxx |
| Cigarettes (including roll-ups) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Cigars | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Tobacco (e.g. pipe) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Others (e.g. nicotine patches, chewing | XX | XX | XX | XX | XX | |
| tobacco) | | | | | | |
| Missing | | | | | | |

<sup>-</sup> The last available assessment before or at date of start of study treatment is taken as "baseline" assessment.

<sup>-</sup> Body mass index (kg/m2): very severely underweight (less than 15.0), severely underweight (>=15.0-<=16.0), underweight (>16.0-<=18.5), normal (>18.5-<=25.0), overweight (>25.0-<=30.0), obese class I (>30.0-<=35.0), obese class II (>35.0-<=40.0) and obese class III (over 40.0).

<sup>-</sup> Time since stopped smoking = (date of screening visit - date stopped smoking + 1) / 30.4375.

<sup>-</sup> Percentage based on the number of patients included in the analysis population (N).

<sup>\$</sup> Comparison Randomized vs Not Randomized. # P-value: For categorical variables Pearson Chi-square test or Fisher's exact test depending on the crosstabulation frequencies. For numeric variables independent t-test for means, Median test for medians. \* p-value<0.05, \*\* p-value<0.01.

#### << Programming note:

Comparison between Randomized and No Randomized group will be done for Demographics and baseline characteristics, History of prior Imatinib therapy, Cardiovascular risk factors, using: Pearson's Chi-square test p-value, or Fisher's exact test in case we have one or more frequencies in the cross-tabulation MR4.0 Yes/No\*Randomized/Not Randomized, less than 5 for categorical variables, to check correlation between MR4.0 and Randomization group.

For numeric variables, Independent t-test for means (using "Equal" variances or "Unequal" variances depending on Variance test result) and Median test for median will be used to test for differences between Randomized and Not Randomized group.

-Pearson's Chi-square test p-value will be the first choice for categorical variables.

Fisher's exact test will be used in case we have one or more frequencies in the cross-tabulation Variable\*Randomized/Not Randomized, less than 5. >>

### Table 14.1-3.1.1 Demographic and characteristics at baseline LSC sub-study Full Analysis Set

<< Programming note: Same shell as table 14.1-3.1, for LSC sub-study FAS patients >>
#### **Table 14.1-4.1 Disease history – Full Analysis Set**

| Disease history | Arm 1 | Arm 2 | Randomized | Not Randomized | Total |
|---|---|---|---|---|---|
| | N=xx | N=xx | N=xx | N=xx | N=xx |
| Time since initial diagnosis (months) | | | | | |
| n | XXX | XXX | XXX | XXX | XXX |
| Mean | xx.x | XX.X | XX.X | XX.X | XX.X |
| SD | x.xx | X.XX | X.XX | X.XX | X.XX |
| 25th Percentile | XX.X | XX.X | XX.X | XX.X | XX.X |
| Median | xx.x | XX.X | XX.X | XX.X | XX.X |
| 75th Percentile | xx.x | XX.X | XX.X | XX.X | XX.X |
| Min-Max | xx.x- xx.x | xx.x- xx.x | xx.x- xx.x | xx.x- xx.x | xx.x- xx.x |
| Time since initial diagnosis (years) | | | | | |
| - n (%)[1] | n=xx | n=xx | n=xx | n=xx | n=xx |
| <2 years | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2 to 4 years | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 4 to 6 years | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 6 to 8 years | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 8 to 10 years | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 10 to 12 years | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| >= 12 years | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Peripheral blood blasts % at diagnosis | | | | | |
| n | XXX | XXX | XXX | XXX | XXX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | X.XX | X.XX | X.XX | X.XX | X.XX |
| 25th Percentile | XX.X | XX.X | XX.X | XX.X | XX.X |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| 75th Percentile | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min-Max | XX.X- XX.X | xx.x- xx.x | xx.x- xx.x | xx.x- xx.x | xx.x- xx.x |
| PB eosinophils % at diagnosis | | | | | |
| n | xxx | XXX | XXX | XXX | XXX |
| Mean | xx.x | XX.X | XX.X | XX.X | XX.X |
| SD | x.xx | X.XX | X.XX | X.XX | X.XX |
| 25th Percentile | xx.x | XX.X | XX.X | XX.X | XX.X |
| Median | xx.x | XX.X | XX.X | XX.X | XX.X |
| 75th Percentile | XX.X | XX.X | XX.X | XX.X | XX.X |

| Novartis<br>RAP Module 7.1 | Confidential<br>6-May-2021 (14:35) | | | Protocol No CA | Page 168<br>AMN107AIC0 |
|---|---|---|---|---|---|
| Min-Max | xx.x- xx.x | xx.x- xx.x | xx.x- xx.x | xx.x- xx.x | xx.x- xx.x |
| PB basophils % at diagnosis | | | | | |
| n | XXX | XXX | XXX | XXX | XXX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | X.XX | X.XX | X.XX | X.XX | X.XX |
| 25th Percentile | XX.X | XX.X | XX.X | XX.X | XX.X |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| 75th Percentile | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min-Max | xx.x- xx.x | XX.X- | xx.x- xx.x | xx.x- xx.x | xx.x- xx.x |
| Platelets at diagnosis (10E9/L) | | | | | |
| n | XXX | XXX | XXX | XXX | XXX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | x.xx | X.XX | X.XX | X.XX | X.XX |
| 25th Percentile | xx.x | XX.X | XX.X | XX.X | XX.X |
| Median | xx.x | XX.X | XX.X | XX.X | XX.X |
| 75th Percentile | xx.x | XX.X | XX.X | XX.X | XX.X |
| Min-Max | xx.x- xx.x | xx.x- xx.x | xx.x- xx.x | xx.x- xx.x | xx.x- xx.x |
| Spleen size at diagnosis (cm under costal margin) | | | | | |
| n | XXX | XXX | XXX | XXX | XXX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | X.XX | X.XX | X.XX | X.XX | X.XX |
| 25th Percentile | XX.X | XX.X | XX.X | XX.X | XX.X |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| 75th Percentile | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min-Max | xx.x- xx.x | xx.x- xx.x | xx.x- xx.x | xx.x- xx.x | xx.x- xx.x |
| Extramedullary involvement other than hepato and/or splenomegaly | | | | | |
| - n (%)[1] | n=xx | n=xx | n=xx | n=xx | n=xx |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Sokal score | | | | | |
| n | XXX | XXX | xxx | XXX | xxx |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | x.xx | X.XX | X.XX | X.XX | X.XX |
| 25th Percentile | XX.X | XX.X | XX.X | XX.X | XX.X |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| ********* | 2323 + 23 | 2121 • 21 | 2323 * 23 | 2323 • 23 | 2121 • 21 |

| Novartis RAP Module 7.1 | Confidential<br>6-May-2021 (14:35) | | | | Page 169<br>Protocol No CAMN107AIC0 |
|---|---|---|---|---|---|
| 75th Percentile<br>Min-Max | xx.x<br>xx.x- xx.x | xx.x<br>xx.x- xx.x | xx.x<br>xx.x- xx.x | xx.x<br>xx.x- xx.x | xx.x<br>xx.x- xx.x |
| - n (%)[1]<br>Low risk | n=xx<br>xx (xx.x) | n=xx<br>xx (xx.x) | n=xx<br>xx (xx.x) | n=xx<br>xx (xx.x) | n=xx<br>xx (xx.x) |
| High risk | xx (xx.x)<br>xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x)<br>xx (xx.x) |
| Euro (Hasford) score | | | | | |
| n | XXX | XXX | XXX | XXX | XXX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | X.XX | X.XX | X.XX | X.XX | X.XX |
| 25th Percentile | XX.X | XX.X | XX.X | XX.X | XX.X |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| 75th Percentile | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min-Max | xx.x- xx.x | xx.x- xx.x | xx.x- xx.x | xx.x- xx.x | xx.x- xx.x |
| - n (%)[1] | n=xx | n=xx | n=xx | n=xx | n=xx |
| Low risk | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Intermediate risk | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| High risk | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| EUTOS score | | | | | |
| n | XXX | XXX | XXX | XXX | XXX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | x.xx | X.XX | X.XX | X.XX | X.XX |
| 25th Percentile | XX.X | XX.X | XX.X | XX.X | XX.X |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| 75th Percentile | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min-Max | xx.x- xx.x | xx.x- xx.x | xx.x- xx.x | xx.x- xx.x | xx.x- xx.x |
| - n (%)[1] | n=xx | n=xx | n=xx | n=xx | n=xx |
| Low risk | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| High risk | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Previous progression to AP/BC | | | | | |
| - n (%)[1] | n=xx | n=xx | n=xx | n=xx | n=xx |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

| Novartis<br>RAP Module 7.1 | Confidential<br>6-May-2021 (14:35 | 5) | | Protocol No | Page 170<br>CAMN107AIC0 |
|---|---|---|---|---|---|
| | vy (- 100 c | • ) | | | |
| Attempt to stop treatment with Imatinib | n=xx | n=xx | n=xx | n=xx | n=xx |
| - n (%)[1] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | | | | | |
| BCR-ABL(IS) ratio at screening | n=xx | n=xx | n=xx | n=xx | n=xx |
| - n (%)[1] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| BCR-ABL(IS) >1% | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| BCR-ABL(IS) >0.1% - <= 1% | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| BCR-ABL(IS) >0.01% - <= 0.1% | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| BCR-ABL(IS) <=0.01% | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Undetectable BCR-ABL | | | | | |
| BCR-ABL(IS) ratio at Re-screening | n=xx | n=xx | n=xx | n=xx | n=xx |
| - n (%)[1] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| BCR-ABL(IS) >1% | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| BCR-ABL(IS) >0.1% - <= 1% | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| BCR-ABL(IS) >0.01% - <= 0.1% | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| BCR-ABL(IS) <=0.01% | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Undetectable BCR-ABL | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

<sup>-</sup> Time since initial diagnosis =  $(date \ of \ the \ baseline \ visit - \ date \ of \ initial \ diagnosis)/30.4375.$ 

#### Table 14.1-4.1.1 Disease history – LSC sub-study Full Analysis Set

<< Programming note: Same shell as table 14.1-4.1, for LSC sub-study FAS patients >>

<sup>-</sup> Sokal score: low risk (<0.8), intermediate risk (>=0.8-<=1.2) and high risk (>1.2).

<sup>-</sup> Euro (Hasford) score: low risk (<=780), intermediate risk (>780-<=1480) and high risk (>1480).

<sup>-</sup> EUTOS score: low risk (<=87) and high risk (>87).

<sup>[1]</sup> Percentages over Number of non-missing.

Table 14.1-5.1 History of prior Imatinib therapy – Full Analysis Set

| | Arm 1<br>N=xx | Arm 2<br>N=xx | Randomized<br>N=xx | Not Randomized<br>N=xx | Total<br>N=xx | Comparison\$<br>p-value# |
|---|---|---|---|---|---|---|
| Prior imatinib intake - n (%) | | | | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | 0.xxx |
| Missing | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Duration of prior exposure (years) | | | | | | |
| - n (%)[1] | n=xx | n=xx | n=xx | n=xx | n=xx | |
| <2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | 0.xxx* |
| >=2 - <5 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| >=5 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Duration of prior exposure (months) | | | | | | |
| n | XXX | XXX | XXX | XXX | XXX | 0.xxx |
| Mean | XX.X | XX.X | XX.X | xx.x | XX.X | 0.xxx |
| SD | XX.XX | XX.XX | XX.XX | xx.xx | XX.XX | |
| 25th Percentile | XX.X | XX.X | XX.X | xx.x | XX.X | |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | |
| 75th Percentile | XX.X | XX.X | XX.X | XX.X | xx.x | |
| Min-Max | xx.x- xx.x | xx.x- xx.x | xx.x- xx.x | xx.x- xx.x | xx.x- xx.x | |

<sup>-</sup> Imatinib therapy starting before the date of first Nilotinib intake.

<sup>-</sup> Duration of prior exposure (months) = (end date of prior imatinib intake - start date of prior imatinib intake + 1)/30.4375.

<sup>- [1]</sup> Percentages based on the number of patients from the analysis population without missing data (n).

<sup>\$</sup> Comparison Randomized vs Not Randomized.

<sup>#</sup> p-value: For categorical variables Pearson Chi-square test or Fisher's exact test depending on the crosstabulation frequencies. For numeric variables independent t-test for mean, Median test for medians.

<sup>\*</sup> p-value<0.05, \*\* p-value<0.01.

#### << Programming note:

Comparison between Randomized and No Randomized group will be done for Demographics and baseline characteristics, History of prior Imatinib therapy, Cardiovascular risk factors, using: Pearson's Chi-square test p-value, or Fisher's exact test in case we have one or more frequencies in the cross-tabulation MR4.0 Yes/No\*Randomized/Not Randomized, less than 5 for categorical variables, to check correlation between MR4.0 and Randomization group.

For numeric variables, Independent t-test for means (using "Equal" variances or "Unequal" variances depending on Variance test result) and Median test for median will be used to test for differences between Randomized and Not Randomized group.

-Pearson's Chi-square test p-value will be the first choice for categorical variables.

Fisher's exact test will be used in case we have one or more frequencies in the cross-tabulation Variable\*Randomized/Not Randomized, less than 5. >>

#### Table 14.1-5.1.1 History of prior Imatinib therapy – LSC sub-study Full Analysis Set

<< Programming note: Same shell as table 14.1-5.1, for LSC sub-study FAS patients >>

Table 14.1-5.2 Prior antineoplastic therapy, other than Imatinib, by ATC class and preferred term - Full Analysis Set

| | Arm 1<br>N=xx<br>n (%) | Arm 2<br>N=xx<br>n (%) | Randomized N=xx n (%) | Not Randomized<br>N=xx<br>n (%) | Total<br>N=xx<br>n (%) |
|---|---|---|---|---|---|
| Any ATC class<br>-Total | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ATC class 1 -Total Preferred term 1 Preferred term 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ATC class 2 -Total Preferred term 1 Preferred term 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

<sup>-</sup> ATC classes are presented alphabetically; preferred terms are sorted within ATC class by descending frequency.

<sup>-</sup> A medication can appear with more than one ATC class.

#### Table 14.1-6.1 Cardiovascular risk factors at baseline – Full Analysis Set

| Cardiovascular factors | Arm 1<br>N=xx | Arm 2<br>N=xx | Randomized<br>N=xx | Not Randomized N=xx | Total<br>N=xx | Comparison\$<br>p-value# |
|---|---|---|---|---|---|---|
| CV risk factor - n (%)[1] | n=xx | n=xx | n=xx | n=xx | n=xx | |
| Very high risk | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | 0.xxx* |
| High risk | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Moderate risk | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Low risk | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |

<sup>-</sup> CV risk factors are defined as described in European Guidelines on cardiovascular disease prevention in clinical practice (version 2012). European Heart Journal (2012) 33, 1635-1701.

#### << Programming note:

Comparison between Randomized and No Randomized group will be done for Demographics and baseline characteristics, History of prior Imatinib therapy, Cardiovascular risk factors, using: Pearson's Chi-square test p-value, or Fisher's exact test in case we have one or more frequencies in the cross-tabulation MR4.0 Yes/No\*Randomized/Not Randomized, less than 5 for categorical variables, to check correlation between MR4.0 and Randomization group.

For numeric variables, Independent t-test for means (using "Equal" variances or "Unequal" variances depending on Variance test result) and Median test for median will be used to test for differences between Randomized and Not Randomized group.

-Pearson's Chi-square test p-value will be the first choice for categorical variables.

Fisher's exact test will be used in case we have one or more frequencies in the cross-tabulation Variable\*Randomized/Not Randomized, less than 5. >>

<sup>- [1]</sup> Percentages over Number of non-missing.

<sup>\$</sup> Comparison Randomized vs Not Randomized.

<sup>#</sup> P-value: For categorical variables Pearson Chi-square test or Fisher's exact test depending on the crosstabulation frequencies.

<sup>\*</sup> p-value<0.05, \*\* p-value<0.01.

# Table 14.1-6.2 Cardiovascular risk factors (based on medical history, laboratory values and vital signs at baseline) – Full Analysis Set Arm 1 Arm 2 Randomized Not Randomized Total

| | Arm 1<br>N=xx | Arm 2<br>N=xx | Randomized<br>N=xx | Not Randomized N=xx | Total<br>N=xx |
|---|---|---|---|---|---|
| Cardiovascular<br>Characteristic | | | | | |
| Medical history - n (%) | | | | | |
| CVEs (IHD: Ischemic heart disease) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| CVEs (PAOD: Peripheral arterial occlusive disease) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| CVEs (ICE: Ischemic cerebrovascular events) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| CVEs (Others) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Hypercholesterolemia | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Hypertension | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Diabetes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| At least one CV medical history | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Fasting glucose at baseline - n (%) | n=xx | n=xx | n=xx | n=xx | n=xx |
| 5.6 - 6.9 mmol/L | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| > 6.9 mmol/L | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Total cholesterol at baseline - n (%) | n=xx | n=xx | n=xx | n=xx | n=xx |
| > 5.2 mmol/L | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| LDL cholesterol at baseline - n (%) | n=xx | n=xx | n=xx | n=xx | n=xx |
| > 3.3 mmol/L | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| HDL cholesterol at baseline - n (%) | n=xx | n=xx | n=xx | n=xx | n=xx |
| <1.3 mmol/L | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Triglycerides at baseline - n (%) | n=xx | n=xx | n=xx | n=xx | n=xx |
| > 1.7 mmol/L | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Total cholesterol, LDL, triglycerides and HDL at baseline - n (%) $^{\star}$ | n=xx | n=xx | n=xx | U=XX | n=xx |
| At least one risk factor** | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

|----------------|--------------------|-------------------------|
| RAP Module 7.1 | 6-May-2021 (14:35) | Protocol No CAMN107AIC0 |

| Blood pressure at baseline - n (%)> 140/90 mmHg | u=xx | n=xx | n=xx | n=xx | n=xx |
|---|---|---|---|---|---|
| Overall Of patient in post-randomization consolidation phase (Arm 2) | xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>NA | xx (xx.x)<br>xx (xx.x) |
| Of patient in TFR phase Of patient in re-treatment phase | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | NA<br>NA | xx (xx.x)<br>xx (xx.x) |

<sup>-</sup> The last available assessment before or at date of start of study treatment is taken as "baseline" assessment.

<sup>-</sup> Blood pressure at baseline (systolic blood pressure > 140mmHg or diastolic blood pressure >90 mmHg).

<sup>\*</sup> number of patients with at least one observation available for total cholesterol, LDL, triglycerides and HDL.

<sup>\*\*</sup> number of patients with high total cholesterol, high LDL, high triglycerides or low HDL.

<sup>-</sup> Percentage based on the number of patients without missing data included in the analysis population (N).

Section 14.2 – Efficacy and other non-safety data (e.g. PK, PK/PD, Health Econ., QoL)

Figures (Section 14.2)

Figure 14.2-1.1 Box-plot of BCR-ABL ratio (IS) during pre-randomization Induction/Consolidation phase – Full Analysis Set



Time-points over Induction/Consolidation phase

- The last value of BCR-ABL (IS) ratio per time-window is displayed in this figure.

- Continue for Arm 2, Not Randomized.
- Display LTWBCRIS values on a logarithmic at base 10 scale (after excluding null value)
- Header/title/footer of the figure must not be displayed in the header and footer of the .doc files >>;

### Figure 14.2-1.2 Box-plot of BCR-ABL ratio (IS) during post-randomization Consolidation phase (ARM 2) – Subset of Full Analysis Set randomized to ARM 2

<< Programming note:

-Same shell as Box-plot of BCR-ABL ratio (IS) during pre-randomization Induction/Consolidation phase - All treated patients (Figure 14.2-1.1) but only for ARM 2, using x-axis label 'Time-points over post-randomization Consolidation phase (ARM2)' and Months 27, 30, 33 and 36 as axis points.

No need to present Baseline.

#### Figure 14.2-1.3 Box-plot of BCR-ABL ratio (IS) during TFR phase – Subset of Full Analysis Set entered TFR

<< Programming note:

-Same shell as Box-plot of BCR-ABL ratio (IS) during pre-randomization Induction/Consolidation phase - All treated patients (Figure 14.2-1.1) but for TFR period, using x-axis label 'Time-points over TFR phase'.

Axis tick points:

Arm1: Month 1, Month 2, Month 3, Month 4, Month 5, Month 6, Month 8, Month 10, Month 12, Month 15, then every 3 months until Month 36.

Arm2: Month 1, Month 2, Month 3, Month 4, Month 5, Month 6, Month 8, Month 10, Month 12, Month 15, then every 3 months until Month 24.

No need to present Baseline.

#### Figure 14.2-1.4 Box-plot of BCR-ABL ratio (IS) during re-treatment phase – Subset of Full Analysis Set entered re-treatment

<< Programming note:

-Same shell as Box-plot of BCR-ABL ratio (IS) during pre-randomization Induction/Consolidation phase - All treated patients (Figure 14.2-1.1) but for re-treatment period, using x-axis label 'Time-points over Re-treatment phase'.

Axis tick points:

Arm1: Day 1, Week 6, Month 3, Month 6, then every 3 months until M36 Arm2: Day 1, Week 6, Month 3, Month 6, then every 3 months until M24 No need to present Baseline.

#### Figure 14.2-1.5 Box-plot of BCR-ABL ratio (IS) during TFR phase – , SDV sensitivity Subset of Full Analysis Set entered TFR

<< Programming note: Same shell as Figure 14.2-1.3, for SDV sensitivity analysis>>
Add footnote:

- SDV sensitivity: Excluding patient visits involved in SDV issues during final data review due to COVID-19.

#### Figure 14.2-1.6 Box-plot of BCR-ABL ratio (IS) during re-treatment phase, SDV sensitivity —Subset of Full Analysis Set entered re-treatment

<< Programming note: Same shell as Figure 14.2-1.4, for SDV sensitivity analysis>> Add footnote:

- SDV sensitivity: Excluding patient visits involved in SDV issues during final data review due to COVID-19.

Figure 14.2-2.1.1 Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase - Full Analysis Set



Figure 14.2-2.1.2 Raw cumulative incidence of MMR during post-randomization Consolidation phase (ARM 2) - Subset of Full Analysis Set randomized to ARM 2

<<Pre><<Pre>rogramming note:

-Same shell as Raw cumulative incidence of MMR during Induction/Consolidation phase (Figure 14.2-2.1.1) but for ARM 2 patients only.>> Axis title: "Time since study start (months)" and Months 27, 30, 33, 36 as axis points

<sup>&</sup>lt;< Programming note:

<sup>-</sup> Display up to Month 24

<sup>-</sup> Header/title/footer of the figure must not be displayed in the header and footer of the .doc files , and Months 0, 3,..., 24 as axis points

## Figure 14.2-2.2.1 Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase by halving time of BCR-ABL (IS) ratio - Full Analysis Set

<< Programming note:

-Same shell as Raw cumulative incidence of MMR during Induction/Consolidation phase (Figure 14.2-2.1.1) but done by subgroup of halving time of BCR-ABL (IS) ratio.>>

#### Figure 14.2-2.2.2 Raw cumulative incidence of MMR during post-randomization Consolidation phase (ARM 2) by halving time of BCR-ABL (IS) ratio - Subset of Full Analysis Set randomized to ARM 2

<< Programming note:

-Same shell as Raw cumulative incidence of MMR during post-randomization consolidation phase (Figure 14.2-2.1.2) but done by subgroup of halving time of BCR-ABL (IS) ratio.>>

# Figure 14.2-2.3.1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase – Full Analysis Set

<< Programming note:

-Same shell as Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase (Figure 14.2-2.1.1) done for MR 4.0.>>

#### Figure 14.2-2.3.2 Raw cumulative incidence of MR 4.0 during post-randomization Consolidation phase (ARM 2) - Subset of Full Analysis Set randomized to ARM 2

<< Programming note:

-Same shell as Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase (Figure 14.2-2.3.1) done for ARM 2 patients only.>>

NovartisConfidentialPage 184RAP Module 7.16-May-2021 (14:35)Protocol No CAMN107AIC0

Figure 14.2-2.3.11 Raw cumulative incidence of MR 4.0, Randomized vs Not Randomized, during prerandomization Induction/Consolidation phase - Full Analysis Set



Figure 14.2-2.4.1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase by halving time of BCR-ABL (IS) ratio - Full Analysis Set

<<Pre><<Pre>rogramming note:

<sup>-</sup>Same shell as Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase by halving time of BCR-ABL (IS) ratio (Figure 14.2-2.2.1) done for MR 4.0.>>

### Figure 14.2-2.4.2 Raw cumulative incidence of MR 4.0 during post-randomization Consolidation phase (ARM 2) by halving time of BCR-ABL (IS) ratio - Subset of Full Analysis Set randomized to ARM 2

<<pre><<Pre>rogramming note:

-Same shell as Raw cumulative incidence of MMR during Induction/Consolidation phase (Figure 14.2-2.4.1) but for ARM 2 patients only.>>

### Figure 14.2-2.5.1 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase - Full Analysis Set

<< Programming note:

-Same shell as Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase (Figure 14.2-2.1.1) done for MR 4.5.>>

#### Figure 14.2-2.5.11 Raw cumulative incidence of MR 4.5, Randomized vs Not Randomized, during prerandomization Induction/Consolidation phase- Full Analysis Set

<<pre><<Programming note: -Same shell as Raw Cumulative incidence of MR 4.0, Randomized vs Not Randomized, during pre-randomization
Induction/Consolidation phase, All treated patients (Figure 14.2-2.3.11), but for MR 4.5.</pre>

#### Figure 14.2-2.5.2 Raw cumulative incidence of MR 4.5 during post-randomization Consolidation phase (ARM 2) - Subset of Full Analysis Set randomized to ARM 2

<< Programming note:

-Same shell as Raw cumulative incidence of MMR during post-randomization Consolidation phase (ARM 2) (Figure 14.2-2.1.1) done for MR 4.5.>>

#### Figure 14.2-2.6.1 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase by halving time of BCR-ABL (IS) ratio - Full Analysis Set

<< Programming note:

-Same shell as Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase by halving time of BCR-ABL (IS) ratio (Figure 14.2-2.2.1) done for MR 4.5 by subgroup of halving time of BCR-ABL (IS) ratio.>>

#### Figure 14.2-2.6.2 Raw cumulative incidence of MR 4.5 during post-randomization Consolidation phase (ARM 2) by halving time of BCR-ABL (IS) ratio - Subset of Full Analysis Set randomized to ARM 2

<< Programming note:

-Same shell as Raw cumulative incidence of MMR during post-randomization Consolidation phase (ARM 2) by halving time of BCR-ABL (IS) ratio - Subgroup of All treated patients randomized to ARM 2 (Figure 14.2-2.2.2) done for MR 4.5 >>

# Figure 14.2-2.7.1 Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase - Full Analysis Set patients not reaching MMR at baseline

<< Programming note:

-Same shell as Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase (Figure 14.2-2.1.1), performed on the subset of subjects not reaching MMR at baseline (i.e. time-to-first MMR not equal to 0). >>

# Figure 14.2-2.8.1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase - Full Analysis Set patients not reaching MR 4.0 at baseline

<< Programming note:

-Same shell as Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase (Figure 14.2-2.1.1), performed on the subset of subjects not reaching MR 4.0 at baseline (i.e. time-to-first MR 4.0 not equal to 0). >>

#### Figure 14.2-2.9.1 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase - Full Analysis Set patients not reaching MR 4.5 at baseline

<< Programming note:

-Same shell as Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase (Figure 14.2-2.1.1), performed on the subset of subjects not reaching MR 4.5 at baseline (i.e. time-to-first MR 4.5 not equal to 0). >>

# Figure 14.2-2.9.2 Raw cumulative incidence of MR 4.5 during post-randomization Induction/Consolidation phase (ARM 2)- Subset of Full Analysis Set patients not reaching MR 4.5 at baseline, randomized to ARM 2.

<< Programming note:

-Same shell as Raw cumulative incidence of MR 4.5 during post-randomization Consolidation phase (ARM 2) (Figure 14.2-2.1.2) performed on the subset of subjects not reaching MR 4.5 at baseline (i.e. time-to-first MR 4.0 not equal to 0). >>

Figure 14.2-2.10.1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase by BCR-ABL(IS) ratio at baseline - Full Analysis Set



<< Programming note:

Continue for Arm 2, Not Randomized.

Figure 14.2-2.10.2 Raw cumulative incidence of MR 4.0 during post-randomization Consolidation phase (ARM 2) by BCR-ABL(IS) ratio at baseline - Subset of Full Analysis Set randomized to ARM 2.

<sup>-</sup> Same shell as Figure 4.4 made by BCR-ABL(IS) ratio (use MRCATBL = 2 for BCR-ABL(IS) ratio >0.1% -  $\le1\%$ , and MRCATBL = 3 for BCR-ABL(IS) ratio >0.01% -  $\le0.1\%$ )

<sup>-</sup> Header/title/footer of the figure must not be displayed in the header and footer of the .doc files >>

<sup>-</sup> Same shell as Figure 14.2-2.10.1, but for ARM 2 patients only.

<sup>-</sup> Header/title/footer of the figure must not be displayed in the header and footer of the .doc files >>

### Figure 14.2-2.11.1 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase by BCR-ABL(IS) ratio at baseline - Full Analysis Set

<< Programming note:

- Same shell as Figure 14.2-2.10.1, but on MR 4.5
- Header/title/footer of the figure must not be displayed in the header and footer of the .doc files >>

#### Figure 14.2-2.11.2 Raw cumulative incidence of MR 4.5 during post-randomization Consolidation phase (ARM 2) by BCR-ABL(IS) ratio at baseline - Subset of Full Analysis Set randomized to ARM 2.

- Same shell as Figure 14.2-2.10.2, but on MR 4.5
- Header/title/footer of the figure must not be displayed in the header and footer of the .doc files >>

Figure 14.2-2.12.1 Box-plot of BCR-ABL ratio (IS) during pre-randomization Induction/Consolidation phase, excluding outliers (BCR-ABL (IS) ratio>10 - Full Analysis Set



- The last value of BCR-ABL (IS) ratio per time-window is displayed in this figure.

#### << Programming note:

- Continue for Arm 2, Not Randomized.
- Same shell as Figure 4.1 but without outliers
- Add footnote "Outliers with BCR-ABL (IS) ratio higher than 10 are not displayed on this figure.>>

Figure 14.2-2.12.2 Box-plot of BCR-ABL ratio (IS) over post-randomization Consolidation phase (ARM 2), excluding outliers (BCR-ABL (IS) ratio>10 - Subset of Full Analysis Set randomized to ARM 2.

<sup>-</sup> Same shell as Figure 14.2-2.12.1, only for ARM 2.

<sup>-</sup> Header/title/footer of the figure must not be displayed in the header and footer of the .doc files >> No need to present Baseline.

# Figure 14.2-2.12.3 Overall box-plot of BCR-ABL ratio (IS) during pre-randomization Induction/Consolidation phase – Full Analysis Set

- X Axis should include: Baseline, Month 3, Month 6,..., Month 24 »»
- X axis label : month

Figure 14.2-13.1 Raw cumulative incidence of loss of MMR during TFR – Subset of Full Analysis Set entering the TFR phase



<< Programming note:

Label of axis to change with: "Time since start of TFR phase (months)" >>

- Axis should go from 0 to month 36
- Graph should be presented using 2 different type of lines ARM 1 (dash) / ARM 2 (full line)

## Figure 14.2-13.2 Raw cumulative incidence of MMR during re-treatment phase – Subset of Full Analysis Set entering the re-treatment phase

<< Programming note: same shell as figure 14.2-13.1 "Time since start of Re-treatment phase (months)" >>

- Axis should go from 0 to month 36 >>>>

### Figure 14.2-13.3 Raw cumulative incidence of loss of MMR during TFR, SDV sensitivity – Subset of Full Analysis Set entering the TFR phase

<< Programming note: Same shell as Figure 14.2-13.1, for SDV sensitivity analysis>>
Add footnote:
- SDV sensitivity: Excluding patient visits involved in SDV issues during final data review due to COVID-19.

#### Figure 14.2-13.4 Raw cumulative incidence of MMR during re-treatment phase, SDV sensitivity – Subset of Full Analysis Set entering the re-treatment phase

<< Programming note: Same shell as Figure 14.2-13.2, for SDV sensitivity analysis>>
Add footnote:
- SDV sensitivity: Excluding patient visits involved in SDV issues during final data review due to COVID-19.

#### Figure 14.2-14.1 Raw cumulative incidence of loss of MR4.0 during TFR phase –Subset of Full Analysis Set entering the TFR phase

- << Programming note: same shell as figure 14.2-13.1 but for TFR MR4.0.
  - Label of axis to change with: "Time since start of TFR phase (months)" >>

# Figure 14.2-14.2 Raw cumulative incidence of MR4.0 during re-treatment phase – Subset of Full Analysis Set entering the re-treatment phase

<< Programming note: same shell as figure 14.2-13.2, but for re-treatment MR4.0 >>

# Figure 14.2-14.3 Raw cumulative incidence of loss of MR4.0 during TFR phase, SDV sensitivity –Subset of Full Analysis Set entering the TFR phase

<< Programming note: Same shell as Figure 14.2-14.1, for SDV sensitivity analysis>>
Add footnote:

- SDV sensitivity: Excluding patient visits involved in SDV issues during final data review due to COVID-19.

# Figure 14.2-14.4 Raw cumulative incidence of MR4.0 during re-treatment phase, SDV sensitivity – Subset of Full Analysis Set entering the re-treatment phase

<< Programming note: Same shell as Figure 14.2-14.2, for SDV sensitivity analysis>>
Add footnote:

- SDV sensitivity: Excluding patient visits involved in SDV issues during final data review due to COVID-19.

#### Figure 14.2-15.1 Raw cumulative incidence of loss of MR4.5 during TFR phase – Subset of Full Analysis Set entering the TFR phase with MR4.5

<< Programming note: same shell as figure 14.2-13.1 but for TFR MR4.5>>

### Figure 14.2-15.2 Raw cumulative incidence of MR4.5 during re-treatment phase – Subset of Full Analysis Set entering the re-treatment phase

<< Programming note: same shell as figure 14.2-13.2 but for re-treatment MR4.5>>

### Figure 14.2-15.3 Raw cumulative incidence of loss of MR4.5 during TFR phase, SDV sensitivity – Subset of Full Analysis Set entering the TFR phase with MR4.5

<< Programming note: Same shell as Figure 14.2-15.1, for SDV sensitivity analysis>> Add footnote:

- SDV sensitivity: Excluding patient visits involved in SDV issues during final data review due to COVID-19.

### Figure 14.2-15.4 Raw cumulative incidence of MR4.5 during re-treatment phase, SDV sensitivity – Subset of Full Analysis Set entering the re-treatment phase

<< Programming note: Same shell as Figure 14.2-15.2, for SDV sensitivity analysis>>
Add footnote:

- SDV sensitivity: Excluding patient visits involved in SDV issues during final data review due to COVID-19.

Figure 14.2-16 Bar plot MR4.0 at 12 months of TFR phase –Subset of Full Analysis Set entering the TFR phase



Programming Note: Use black color but different patterns for each bar.

Figure 14.2-16.2 Bar plot MR4.0 at month 12 TFR phase , SDV sensitivity –Subset of Full Analysis Set entering the TFR phase

<< Programming note: Same shell as Figure 14.2-16, for SDV sensitivity analysis>>
Add footnote:

<sup>-</sup> SDV sensitivity: Excluding patient visits involved in SDV issues during final data review due to COVID-19.

Figure 14.2-17.1 Kaplan-Meier analysis of progression-free survival during the TFR phase –Subset of Full Analysis Set entering the TFR phase



The axis label should "Time since start of TFR phase (months)"

Months 0-36 for Arm 1, Months 0-24 for Arm 2

Vertical (Y-Axis) label "Prop. of pts. without Disease progression"

Figure 14.2-17.2 Kaplan-Meier analysis of treatment-free survival during the TFR phase –Subset of Full Analysis Set entering the TFR phase

<< Programming note: same shell as figure 14.2-17.1 for TFR treatment free survival
Vertical (Y-Axis) label "Prop. of pts. without treatment">>>

#### Figure 14.2-17.3 Kaplan-Meier analysis of progression-free survival during the TFR phase, SDV sensitivity – Subset of Full Analysis Set entering the TFR phase

<< Programming note: Same shell as Figure 14.2-17.1, for SDV sensitivity analysis>>
Add footnote:

- SDV sensitivity: Excluding patient visits involved in SDV issues during final data review due to COVID-19.

# Figure 14.2-17.4 Kaplan-Meier analysis of treatment-free survival during the TFR phase, SDV sensitivity – Subset of Full Analysis Set entering the TFR phase

<< Programming note: Same shell as Figure 14.2-17.2, for SDV sensitivity analysis>>
Add footnote:

- SDV sensitivity: Excluding patient visits involved in SDV issues during final data review due to COVID-19.

#### Figure 14.2-18.1 Kaplan-Meier analysis of reachievement of MMR, after loss of response in TFR –Subset of Full Analysis Set entering the re-treatment phase

<< Programming note: same shell as figure 14.2-4.1 for re-treatment
Months 0-36 for Arm 1, Months 0-24 for Arm 2
Vertical (Y-Axis) label "Prop. of pts. without re-achievement of MMR">>

#### Figure 14.2-18.2 Kaplan-Meier analysis of reachievement of MR4.0, after loss of response in TFR – Subset of Full Analysis Set entering the re-treatment phase

<< Programming note: same shell as figure 14.2-4.1 for re-treatment
Months 0-36 for Arm 1, Months 0-24 for Arm 2>>
Vertical (Y-Axis) label "Prop. of pts. without re-achievement of MR4.0"

# Figure 14.2-18.3 Kaplan-Meier analysis of reachievement of MMR, after loss of response in TFR, SDV sensitivity —Subset of Full Analysis Set entering the re-treatment phase

<< Programming note: Same shell as Figure 14.2-18.1, for SDV sensitivity analysis>>
Add footnote:

- SDV sensitivity: Excluding patient visits involved in SDV issues during final data review due to COVID-19.

#### Figure 14.2-18.4 Kaplan-Meier analysis of reachievement of MR4.0, after loss of response in TFR, SDV sensitivity – Subset of Full Analysis Set entering the re-treatment phase

<< Programming note: Same shell as Figure 14.2-18.2, for SDV sensitivity analysis>>
Add footnote:

- SDV sensitivity: Excluding patient visits involved in SDV issues during final data review due to COVID-19.

#### Tables (Section 14.2)

Table 14.2-1.1 Description of BCR-ABL (IS) ratio at Month 3 and halving time of BCR-ABL (IS) ratio subgroups – Full Analysis Set

| Subgroups | Arm 1<br>N=xxx<br>n (%) | Arm 2<br>N=xxx<br>n (%) | Randomized<br>N=xxx<br>n (%) | Not Randomized N=xxx n (%) | Total<br>N=xxx<br>n (%) |
|---|---|---|---|---|---|
| BCR-ABL (IS) ratio at Month 3-n (%) <= 0.005% > 0.005% | n=xx | n=xx | n=xx | n=xx | n=xx |
| | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Halving time-n (%) <= 3 months (Day 91) > 3 months (Day 91) | n=xx | n=xx | n=xx | n=xx | n=xx |
| | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

<sup>-</sup> Percentage based on the number of patients with available data (n)

#### Table 14.2-2.1.1 Molecular response MR4.0 at 12 months of TFR-Subset of Full Analysis Set entering the TFR phase

| • | Arm 1 | Arm 2 | Total |
|---|---|---|---|
| | N=xx | N=xx | N=xx |
| Number of responders | xx | xx | xx |
| Percentage (95% CI) | xx (xx.x, xx.x) | xx (xx.x, xx.x) | xx (xx.x, xx.x) |
| Comparison Arm 1 vs Arm 2 p-value\$ | 0.xxx | | |

<sup>-</sup> Responders= Patients still in TFR with >=MR4.0, without molecular relapse.

#### << Programming note:

-The percentage is obtained by dividing the number with response by number of patients entered TFR.>>

Comparison between Randomized and No Randomized group will be done for Demographics and baseline characteristics, History of prior Imatinib therapy, Cardiovascular risk factors, using: Pearson's Chi-square test p-value, or Fisher's exact test in case we have one or more frequencies in the cross-tabulation MR4.0 Yes/No\*Randomized/Not Randomized, less than 5 for categorical variables, to check correlation between MR4.0 and Randomization group.

For numeric variables, Independent t-test for means (using "Equal" variances or "Unequal" variances depending on Variance test result) and Median test for median will be used to test for differences between Randomized and Not Randomized group.

-Pearson's Chi-square test p-value will be the first choice for categorical variables.

Fisher's exact test will be used in case we have one or more frequencies in the cross-tabulation Variable\*Randomized/Not Randomized, less than 5. >>

#### Table 14.2-2.1.2 Molecular response MR4.0 at 12 months of TFR-Subset of Per Protocol Analysis Set entering the TFR phase

<< Programming note: same shell as Table 14.2-2.1.1 for Per Protocol Set

<sup>-</sup> Confidence interval calculated as per Clopper-Pearson exact method.

<sup>-</sup> Percentage based on the number of patients included in the analysis population (N).

<sup>-</sup> Patients entered TFR considered for percentages denominator.

<sup>\$</sup> Pearson Chi-square test or Fisher's exact test depending on the crosstabulation frequencies.

<sup>\*</sup> p-value<0.05, \*\* p-value<0.01.

#### Table 14.2-2.1.3 Molecular response MR4.0 at 12 months of TFR-Full Analysis Set

<< Programming note: same shell as Table 14.2-2.1.1 for Full Analysis Set</pre>

Using the following footnotes:

Responders= Patients still in TFR with >=MR4.0, without molecular relapse.

- Confidence interval calculated as per Clopper-Pearson exact method.
- Percentage based on the number of patients included in the analysis population (N).
- FAS patients considered for percentages denominator.
- Patients randomized to Arm 1 and Arm 2 not entering the TFR phase will be considered as unsuccessful TFR. The same rule described in the previous section will be used to deal with any missing PCR assessment at Month 12.
- \$ Pearson Chi-square test or Fisher's exact test depending on the crosstabulation frequencies.
- \* p-value<0.05, \*\* p-value<0.01.

#### Table 14.2-2.1.4 Molecular response MR4.0 at 12 months of TFR-Per Protocol Analysis Set

<< Programming note: same shell as Table 14.2-2.1.1 for Per Protocol Analysis Set
Using the following footnotes:</pre>

- Responders= Patients still in TFR with >=MR4.0, without molecular relapse.
- Confidence interval calculated as per Clopper-Pearson exact method.
- Percentage based on the number of patients included in the analysis population (N).
- PPS patients considered for percentages denominator.
- Patients randomized to Arm 1 and Arm 2 not entering the TFR phase will be considered as unsuccessful TFR. The same rule described in the previous section will be used to deal with any missing PCR assessment at Month 12.
- \$ Pearson Chi-square test or Fisher's exact test depending on the crosstabulation frequencies.
- \* p-value<0.05, \*\* p-value<0.01.

# Table 14.2-2.1.5 Molecular response MR4.0 at 12 months of TFR- Subset of Full Analysis Set entering the TFR phase with MR4.0 achieved up to month 3 of pre-randomization Induction/Consolidation phase

<< Programming note: same shell as Table 14.2-2.1.1</pre>

# Table 14.2-2.1.6 Molecular response MR4.0 at 12 months of TFR- Subset of Full Analysis Set entering the TFR phase with MR4.5 achieved up to month 3 of pre-randomization Induction/Consolidation phase

<< Programming note: same shell as Table 14.2-2.1.1</pre>

### Table 14.2-2.1.7 Molecular response MR4.0 at 12 months of TFR, SDV sensitivity –Subset of Full Analysis Set entering the TFR phase

<< Programming note: Same shell as Table 14.2-2.1.1, for SDV sensitivity analysis>>
Add footnote:

- SDV sensitivity: Excluding patient visits involved in SDV issues during final data review due to COVID-19.

### Table 14.2-2.1.8 Molecular response MR4.0 at 12 months of TFR, SDV sensitivity –Subset of Per Protocol Analysis Set entering the TFR phase

<< Programming note: Same shell as Table 14.2-2.1.2, for SDV sensitivity analysis>>
Add footnote:

- SDV sensitivity: Excluding patient visits involved in SDV issues during final data review due to COVID-19.

#### Table 14.2-2.1.9 Molecular response MR4.0 at 12 months of TFR, SDV sensitivity –Full Analysis Set

<< Programming note: Same shell as Table 14.2-2.1.3, for SDV sensitivity analysis>>
Add footnote:

- SDV sensitivity: Excluding patient visits involved in SDV issues during final data review due to COVID-19.
#### Table 14.2-2.1.10 Molecular response MR4.0 at 12 months of TFR, SDV sensitivity –Per Protocol Analysis Set

<< Programming note: Same shell as Table 14.2-2.1.4, for SDV sensitivity analysis>> Add footnote:

Table 14.2-2.2.1 Kaplan-Meier analysis of treatment-free survival during the TFR phase – Subset of Full Analysis Set entering the TFR phase

| KM estimates | Arm 1 | Arm 2 |
|---|---|---|
| Number of patients - n(%) | | |
| with events | xx (xx.x) | xx (xx.x) |
| Relapse | xx (xx.x) | xx (xx.x) |
| Re-treatment with Nilotinib | xx (xx.x) | xx (xx.x) |
| Progression to AP-BC | xx (xx.x) | xx (xx.x) |
| Death from any cause | xx (xx.x) | xx (xx.x) |
| Relapse + Death from any cause | xx (xx.x) | xx (xx.x) |
| < <note any="" combinat<="" for="" programming:add="" td=""><td>ion of events occurring on the</td><td>same date&gt;&gt;</td></note> | ion of events occurring on the | same date>> |
| with censorings | xx (xx.x) | xx (xx.x) |
| Time to event (months) | | |
| 25th percentile (95% CI) | xx (xx.x, xx.x) | xx (xx.x xx.x)) |
| Median (95% CI) | xx (xx.x xx.x)) | xx (xx.x xx.x)) |
| 75th percentile (95% CI) | xx (xx.x xx.x)) | xx (xx.x xx.x)) |
| Percentage of patients without event - | | |
| Estimate n(%)(95% CI) | | |
| 6 months | xx (xx.x) (xx.x, xx. | |
| 12 months | xx (xx.x) (xx.x, xx. | x) $xx (xx.x) (xx.x, xx.x)$ |
| 18 months | xx (xx.x) (xx.x, xx. | x) $xx (xx.x) (xx.x, xx.x)$ |
| 24 months | xx (xx.x) (xx.x, xx. | x) $xx (xx.x) (xx.x, xx.x)$ |
| 30 months | xx (xx.x) (xx.x, xx. | x) |
| 36 months | xx (xx.x) (xx.x, xx. | x) |

<sup>-</sup> NE: Not Estimable

<sup>-</sup> Patients randomized to Arm 2 have a maximum of 24 months of TFR phase.

<sup>-</sup> Event = first occurrence of relapse, re-treatment with nilotinib, progression to AP/BC or death for any cause.

<sup>-</sup> Censoring rule = patients who did not meet the event are censored at the first date occurring between: the last contact date, the end of TFR phase and the date of death.

<sup>-</sup> Time to event = (date of event - start date of TFR phase + 1)/30.4375.

<sup>-</sup> n is the number of patients at risk at the timepoint (i.e. without event and still ongoing)

<sup>-</sup> The percentage of patients without event and the respective 95% C.I. are estimated from Kaplan Meier.

#### Table 14.2-2.2.2 Kaplan-Meier analysis of treatment-free survival during the TFR phase – Subset of Per Protocol Analysis Set entering the TFR phase

<< Programming note: same shell as Table 14.2-2.2.1 for Per Protocol Set

#### Table 14.2-2.2.3 Kaplan-Meier analysis of treatment-free survival during the TFR phase, SDV sensitivity – Subset of Full Analysis Set entering the TFR phase

<< Programming note: Same shell as Table 14.2-2.2.1, for SDV sensitivity analysis>>
Add footnote:

- SDV sensitivity: Excluding patient visits involved in SDV issues during final data review due to COVID-19.

#### Table 14.2-2.2.4 Kaplan-Meier analysis of treatment-free survival during the TFR phase, SDV sensitivity – Subset of Per Protocol Analysis Set entering the TFR phase

<< Programming note: Same shell as Table 14.2-2.2.2, for SDV sensitivity analysis>>
Add footnote:

#### Table 14.2-2.3 Kaplan-Meier analysis of overall survival from Randomization-Randomized Set

| KM estimates | Arm 1<br>(N=xxx) | Arm 2 (N=xxx) |
|---|---|---|
| Number of patients - n(%) | | |
| with events (deaths) | xx (xx.x) | xx (xx.x) |
| with censorings | xx (xx.x) | xx (xx.x) |
| Time to event (months) | | |
| 25th percentile (95% CI) | xx (xx.x, xx.x) | xx (xx.x xx.x)) |
| Median (95% CI) | xx (xx.x xx.x)) | xx (xx.x xx.x)) |
| 75th percentile (95% CI) | xx (xx.x xx.x)) | xx (xx.x xx.x)) |
| Percentage of patients without event - Estimate n(%)(95% CI) | | |
| 6 months | xx (xx.x) (xx.x, xx.x) | xx (xx.x) (xx.x, xx.x) |
| 12 months | xx (xx.x) (xx.x, xx.x) | xx (xx.x) (xx.x, xx.x) |
| 18 months | xx (xx.x) (xx.x, xx.x) | xx (xx.x) (xx.x, xx.x) |
| 24 months | xx (xx.x) (xx.x, xx.x) | xx (xx.x) (xx.x, xx.x) |
| 30 months | xx (xx.x) (xx.x, xx.x) | |
| 36 months | xx (xx.x) (xx.x, xx.x) | |

<sup>-</sup> NE: Not Estimable

Event = death for any cause.

<sup>-</sup> Censoring rule = patients who did not meet the event are censored at the first date occurring between: the last contact and the date of death.

<sup>-</sup> Time to event = (date of event - Randomization date + 1)/30.4375.

<sup>-</sup> n is the number of patients at risk at the timepoint (i.e. without event and still ongoing)

<sup>-</sup> The percentage of patients without event and the respective 95% C.I. are estimated from Kaplan Meier.

Table 14.2-2.4 Kaplan-Meier analysis of progression-free survival during the TFR phase — Subset of Full Analysis Set entering the TFR phase

| KM estimates | Arm 1 | Arm 2 |
|---|---|---|
| Number of patients - n(%) | | |
| with events | xx (xx.x) | xx (xx.x) |
| with censorings | xx (xx.x) | xx (xx.x) |
| Time to event (months) | | |
| 25th percentile (95% CI) | xx (xx.x, xx.x) | xx (xx.x xx.x)) |
| Median (95% CI) | xx (xx.x xx.x)) | xx (xx.x xx.x)) |
| 75th percentile (95% CI) | xx (xx.x xx.x)) | xx (xx.x xx.x)) |
| Percentage of patients without event - | | |
| Estimate n(%)(95% CI) | | |
| 6 months | xx (xx.x) (xx.x, xx.x) | xx (xx.x) (xx.x, xx.x) |
| 12 months | xx (xx.x) (xx.x, xx.x) | xx (xx.x) (xx.x, xx.x) |
| 18 months | xx (xx.x) (xx.x, xx.x) | xx (xx.x) (xx.x, xx.x) |
| 24 months | xx (xx.x) (xx.x, xx.x) | xx (xx.x) (xx.x, xx.x) |
| 30 months | xx (xx.x) (xx.x, xx.x) | |
| 36 months | xx (xx.x) (xx.x, xx.x) | |

<sup>-</sup> NE: Not Estimable

<sup>-</sup> Patients randomized to Arm 2 have a maximum of 24 months of TFR phase.

<sup>-</sup> Event = first occurrence of progression to AP/BC or death for any cause.

<sup>-</sup> Censoring rule = patients who did not meet the event are censored at the first date occurring between: the last contact date, the end of TFR phase and the date of death.

<sup>-</sup> Time to event = (date of event - start date of TFR phase + 1)/30.4375.

<sup>-</sup> n is the number of patients at risk at the timepoint (i.e. without event and still ongoing)

<sup>-</sup> The percentage of patients without event and the respective 95% C.I. are estimated from Kaplan Meier.

#### Table 14.2-2.5 Kaplan-Meier analysis of overall survival from Randomization, SDV sensitivity –Randomized Set

<<pre><< Programming note: Same shell as Table 14.2-2.3, for SDV sensitivity analysis>>
Add footnote:

- SDV sensitivity: Excluding patient visits involved in SDV issues during final data review due to COVID-19.

# Table 14.2-2.6 Kaplan-Meier analysis of progression-free survival during the TFR phase, SDV sensitivity — Subset of Full Analysis Set entering the TFR phase

<< Programming note: Same shell as Table 14.2-2.4, for SDV sensitivity analysis>>
Add footnote:

Table 14.2-3.1 Major molecular response during pre-randomization Induction/Consolidation phase –Full Analysis Set

| <b>,</b> | Arm 1<br>N=xx | Arm 2<br>N=xx | Randomized<br>N=xx | Not Randomized<br>N=xx | Total<br>N=xx |
|---|---|---|---|---|---|
| Rate of major molecular response at Baseline Number of responders Response Rate % (95% CI) | xx<br>xx (xx.x, xx.x) | xx<br>xx (xx.x, xx.x) | xx<br>xx (xx.x, xx.x) | xx<br>xx (xx.x, xx.x) | xx<br>xx (xx.x, xx.x) |
| Rate of major molecular response at Month 3 Number of responders Response Rate % (95% CI) | xx<br>xx (xx.x, xx.x) | xx<br>xx (xx.x, xx.x) | xx<br>xx (xx.x, xx.x) | xx<br>xx (xx.x, xx.x) | xx<br>xx (xx.x, xx.x) |
| Rate of major molecular response at Month 6 | | | | | |
| Rate of major molecular response at Month 9 | | | | | |
| Rate of major molecular response at Month 12 | ••• | ••• | ••• | ••• | ••• |
| Rate of major molecular response at Month 15 | | | | | |
| Rate of major molecular response at Month 18 | | | | ••• | |
| Rate of major molecular response at Month 21 | | | | | |
| Rate of major molecular response at Month 24 | ••• | | ••• | ••• | ••• |
| • • • | | | | | |

Rate of major molecular response at Month 24 (Nominal visit\*)

... ... ...

- Rate was computed using time-window as described in the RAP Module 3.
- Percentage based on the number of patients included in the analysis population (N).
- Confidence interval calculated as per Clopper-Pearson exact method.
- \* Nominal visit is according to the CRF record, regardless of time-window derived visit.

#### << Programming note:

- -The number of responders at Month x is obtained by counting all patients with a response on the last assessment of time-window x.
- -The percentage is obtained by dividing the number of responders by N.>>

# Table 14.2-3.1.1 Major molecular response during pre-randomization Induction/Consolidation phase – LSC sub-study Full Analysis Set

<< Programming note: Same shell as table 14.2-3.1, for LSC sub-study FAS>>

Table 14.2-3.2 Major molecular response during post-randomization consolidation phase (ARM 2)– Subset of Full Analysis Set randomized to Arm 2

| | Arm2<br>N=xx |
|---|---|
| Rate of major molecular response at Month 27<br>Number of responders<br>Response Rate % (95% CI) | xx<br>xx (xx.x, xx.x) |
| Rate of major molecular response at Month 27 (Nominal visit*)<br>Number of responders<br>Response Rate % (95% CI) | xx<br>xx (xx.x, xx.x) |
| Rate of major molecular response at Month 30<br>Number of responders<br>Response Rate % (95% CI) | xx<br>xx (xx.x, xx.x) |
| Rate of major molecular response at Month 33 Number of responders | xx |
| Rate of major molecular response at Month 36 | xx<br> |
| Rate of major molecular response at Month 36 (Nominal vist*) | |

<sup>-</sup> Rate was computed using time-window as described in the RAP Module 3.

### Table 14.2-3.2.1 Major molecular response during post-randomization consolidation phase (ARM 2) – LSC substudy Full Analysis Set randomized to Arm 2

<< Programming note: Same shell as table 14.2-3.2, for LSC sub-study FAS ARM 2>>

<sup>-</sup> Percentage based on the number of patients included in the analysis population (N).

<sup>-</sup> Confidence interval calculated as per Clopper-Pearson exact method.

<sup>\*</sup> Nominal visit is according to the CRF record, regardless of time-window derived visit.

Table 14.2-3.3 Major molecular response during TFR phase –Subset of Full Analysis Set patients entered TFR phase

| | Arm 1<br>N=xx | Arm 2<br>N=xx | Total<br>N=xx |
|---|---|---|---|
| Rate of major molecular response at Baseline<br>Number of responders<br>Response Rate % (95% CI) | xx<br>xx (xx.x, xx.x) | xx<br>xx (xx.x, xx.x) | xx<br>xx (xx.x, xx.x) |
| Rate of major molecular response at Month 3<br>Number of responders<br>Response Rate % (95% CI) | xx<br>xx (xx.x, xx.x) | xx<br>xx (xx.x, xx.x) | xx<br>xx (xx.x, xx.x) |
| Rate of major molecular response at Month 6 Rate of major molecular response at Month 9 | | | |
| Rate of major molecular response at Month 12 | | | |
| Rate of major molecular response at Month 15 | | | ••• |
| Rate of major molecular response at Month 18 | | | • • • |
| Rate of major molecular response at Month 21 Rate of major molecular response at Month 24 | ••• | • • • | ••• |
| Rate of major molecular response at Month 24 (Nominal visit*) | | ••• | |
| Rate of major molecular response at Month 27 | ••• | ••• | ••• |
| ••• | • • • | • • • | • • • |

| 6-May-2021 (14:35) | | Protocol No CAMN107AIC0 |
|---|---|---|
| inal visit*) | | |
| ••• | ••• | ••• |
| n 30 | | |
| • • • | • • • | ••• |
| n 33 | | |
| • • • | • • • | ••• |
| n 36 | | |
| • • • | • • • | • • • |
| inal visit*) | | |
| • • • | • • • | ••• |
| | 6-May-2021 (14:35) inal visit*) 1 30 1 33 1 36 inal visit*) | 6-May-2021 (14:35) inal visit*) 1 30 1 33 1 36 inal visit*) |


#### << Programming note:

**Novartis** 

#### Table 14.2-3.4 Major molecular response during re-treatment phase—Subset of Full Analysis Set patients entered re- treatment phase

<< Programming note: Same shell as table 14.2-3.3, time-window: Day 1, Week 6, Month 3 up to Month 36 by 3 for re-treatment two
arms>>

<sup>-</sup> Rate was computed using time-window as described in the RAP Module 3.

<sup>-</sup> Percentage based on the number of patients included in the analysis population (N).

<sup>-</sup> Confidence interval calculated as per Clopper-Pearson exact method.

<sup>\*</sup> Nominal visit is according to the CRF record, regardless of time-window derived visit.

<sup>-</sup>The number of responders at Month x is obtained by counting all patients with a response on the last assessment of time-window x.

<sup>-</sup>The percentage is obtained by dividing the number of responders by N.>>

Table 14.2-3.5 Major molecular response during TFR phase –Subset of Full Analysis Set patients entered TFR phase with MR4.0 achieved up to month 3 of pre-randomization Induction/Consolidation phase

<< Programming note: same shell as Table 14.2-3.3</pre>

Table 14.2-3.6 Major molecular response during TFR phase –Subset of Full Analysis Set patients entered TFR phase with MR4.5 achieved up to month 3 of pre-randomization Induction/Consolidation phase

<< Programming note: same shell as Table 14.2-3.3</pre>

Table 14.2-3.7 Major molecular response during TFR phase, SDV sensitivity –Subset of Full Analysis Set patients entered TFR phase

<< Programming note: Same shell as Table 14.2-3.3, for SDV sensitivity analysis>> Add footnote:

- SDV sensitivity: Excluding patient visits involved in SDV issues during final data review due to COVID-19.

Table 14.2-3.8 Major molecular response during re-treatment phase, SDV sensitivity –Subset of Full Analysis Set patients entered re- treatment phase

<< Programming note: Same shell as Table 14.2-3.4, for SDV sensitivity analysis>>
Add footnote:

#### Table 14.2-4.1 Molecular response 4.0 during pre-randomization Induction/Consolidation phase – Full Analysis Set

<< Programming note: Same shell as table 14.2-3.1, for MR4.0 >>

Table 14.2-4.1.1 Molecular response 4.0 during pre-randomization Induction/Consolidation phase – LSC substudy Full Analysis Set

<< Same shell as table 14.2-3.1, for LSC sub-study FAS MR4.0 ARM 2 >>

Table 14.2-4.2.1 Molecular response 4.0 during post-randomization consolidation phase (ARM 2) – Subset of Full Analysis Set randomized to Arm 2

<< Programming note: Same shell as table 14.2-3.2, for MR4.0 ARM 2>>

Table 14.2-4.2.2 Molecular response 4.0 during post-randomization consolidation phase (ARM 2) – Subset of Per Protocol randomized to Arm 2

<< Programming note: Same shell as table 14.2-4.2.1, for PPS>>
Add footnote:

Per Protocol Analysis Set (PPS) comprises all subjects who are enrolled without major protocol deviation (PD severity codes: 0, 1, 5, 8).

Table 14.2-4.2.11 Molecular response 4.0 during post-randomization consolidation phase (ARM 2) – Subset of LSC sub-study Full Analysis Set randomized to Arm 2

<< Programming note: Same shell as table 14.2-3.1, for LSC sub-study FAS MR4.0 ARM 2>>

#### Table 14.2-4.3.1 Molecular response 4.0 during TFR phase – Subset of Full Analysis Set entering the TFR phase

<< Programming note: Same shell as table 14.2-3.3, for MR4.0 TFR two arms >>

#### Table 14.2-4.3.2 Molecular response 4.0 during TFR phase – Subset of Per Protocol Analysis Set entering the TFR phase

<< Programming note: Same shell as table 14.2-4.3.1, for PPS>>
Add footnote:

Per Protocol Analysis Set (PPS) comprises all subjects who are enrolled without major protocol deviation (PD severity codes: 0, 1, 5, 8).

#### Table 14.2-4.3.3 Molecular response 4.0 during TFR phase, SDV sensitivity – Subset of Full Analysis Set entering the TFR phase

<< Programming note: Same shell as Table 14.2-4.3.1, for SDV sensitivity analysis>>
Add footnote:

Table 14.2-4.4 Molecular response 4.0 during re-treatment phase – Subset of Full Analysis Set entering the retreatment phase

<< Programming note: Same shell as table 14.2-3.4, for MR4.0 re-treatment two arms >>

Table 14.2-4.5 Molecular response 4.0 during TFR phase – Subset of Full Analysis Set entering the TFR phase with MR4.0 achieved up to month 3 of pre-randomization Induction/Consolidation phase

<< Programming note:: same shell as table 14.2-4.3.1 >>

Table 14.2-4.6 Molecular response 4.0 during TFR phase – Subset of Full Analysis Set entering the TFR phase with MR4.5 achieved up to month 3 of pre-randomization Induction/Consolidation phase

<< Programming note: same shell as table 14.2-4.3.1 >>

Table 14.2-4.7 Molecular response 4.0 during re-treatment phase, SDV sensitivity – Subset of Full Analysis Set entering the re-treatment phase

<< Programming note: Same shell as Table 14.2-4.4, for SDV sensitivity analysis>>
Add footnote:

#### Table 14.2-5.1 Molecular response 4.5 during pre-randomization Induction/Consolidation—Full Analysis Set

<< Programming note: Same shell as table 14.2-3.1, for MR4.5, exclude Month 24 (Nominal visit\*) >>

#### Table 14.2-5.1.1 Molecular response 4.5 during pre-randomization Induction/Consolidation— LSC sub-study Full Analysis Set

<< Programming note: Same shell as table 14.2-5.1, for LSC sub-study FAS MR4.5 >>

#### Table 14.2-5.2 Molecular response 4.5 during post-randomization consolidation phase (ARM 2) – Subset of Full Analysis Set randomized to Arm 2

<< Programming note: Same shell as table 14.2-3.2, for MR4.5 ARM 2, exclude Month 27 (Nominal visit\*) and Month 36 (Nominal vist\*)>>

# Table 14.2-5.2.1 Molecular response 4.5 during post-randomization consolidation phase (ARM 2) – Subset of LSC sub-study Full Analysis Set randomized to Arm 2

<< Programming note: Same shell as table 14.2-5.1, for LSC sub-study FAS MR4.5 ARM 2>>

#### Table 14.2-5.3 Molecular response 4.5 during TFR phase – Subset of Full Analysis Set entering the TFR phase

<< Programming note: Same shell as table 14.2-3.3, for MR4.5 TFR two arms, exclude Month 24 (Nominal visit\*), Month 27 (Nominal visit\*) >>

#### Table 14.2-5.4 Molecular response 4.5 during re-treatment phase – Subset of Full Analysis Set entering the retreatment phase

<< Programming note: Same shell as table 14.2-3.4, for MR4.5 re-treatment two arms exclude Month 24 (Nominal visit\*), Month 27
(Nominal visit\*), Month 36 (Nominal visit\*) >>

Table 14.2-5.5 Molecular response 4.5 during TFR phase – Subset of Full Analysis Set entering the TFR phase with MR4.0 achieved up to month 3 of pre-randomization Induction/Consolidation phase

<< Programming note: same shell as table 14.2-5.3 >>

Table 14.2-5.6 Molecular response 4.5 during TFR phase – Subset of Full Analysis Set entering the TFR phase with MR4.5 achieved up to month 3 of pre-randomization Induction/Consolidation phase

<< Programming note: same shell as table 14.2-5.3 >>

#### Table 14.2-5.7 Molecular response 4.5 during TFR phase, SDV sensitivity – Subset of Full Analysis Set entering the TFR phase

<< Programming note: Same shell as Table 14.2-5.3, for SDV sensitivity analysis>>
Add footnote:

- SDV sensitivity: Excluding patient visits involved in SDV issues during final data review due to COVID-19.

#### Table 14.2-5.8 Molecular response 4.5 during re-treatment phase, SDV sensitivity — Subset of Full Analysis Set entering the re-treatment phase

<< Programming note: Same shell as Table 14.2-5.4, for SDV sensitivity analysis>>
Add footnote:

Table 14.2-6.1 Raw cumulative incidence MMR during pre-randomization Induction/Consolidation phase – Full Analysis Set

| | Arm 1 | Arm 2 | Randomized | Not Randomized | Total |
|---|---|---|---|---|---|
| | N=xx | N=xx | N=XX | N=XX | N=xx |
| Major molecular response at baseline | | | | | |
| Number of responders | XX | XX | XX | XX | XX |
| Percentage (95% CI) | xx (xx.x, xx.x) | xx (xx.x, xx.x) | xx (xx.x, xx.x) | xx (xx.x, xx.x) | xx (xx.x, xx.x) |
| Cumulative major molecular response up to 3 months (Day 91) Cumulative number of responders | xx | xx | xx | xx | xx |
| Cumulative percentage (95% CI) | xx (xx.x, xx.x) | xx (xx.x, xx.x) | xx (xx.x, xx.x) | xx (xx.x, xx.x) | xx (xx.x, xx.x) |
| Cumulative major molecular response up to 6 months (Day 183) Cumulative number of responders Cumulative major molecular response up to 9 months (Day | xx<br> | xx<br> | xx<br> | xx<br>··· | xx<br> |
| 274) | | | | | |
| Cumulative major molecular response up to 12 months (Day 365) | | | | | |
| Cumulative major molecular response up to 15 months (Day 457) | ••• | ••• | ••• | ••• | ••• |
| Cumulative major molecular response up to 18 months (Day 548) | ••• | ••• | ••• | ••• | ••• |

| Novartis RAP Module 7.1 | Confidential<br>6-May-2021 (14:35) | | Page 221<br>Protocol No CAMN107AIC0 | |
|---|---|---|---|---|
| Cumulative major molecular response up to2 21 months (Day 639) | ••• | | | ••• |
| Cumulative Major molecular response up to 24 months (Day 731) | | ••• | | |

<sup>-</sup> Percentage based on the number of patients in the analysis population (N).

#### <<pre><<Pre>rogramming note:

-Cumulative number with response at Month x is obtained by counting all patients with a time to response in days before Day x;-The percentage is obtained by dividing the number with response by N.>>

# Table 14.2-6.1.1 Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase – LSC sub-study Full Analysis Set

<< Programming note: Same shell as table 14.2-6.1, for LSC sub-study FAS>>

#### Table 14.2-6.2 Raw cumulative incidence MMR during post-randomization Consolidation phase (ARM 2) - Subset of Full Analysis Set patients randomized to ARM 2

<< Programming note: Same shell as table 14.2-6.1, for ARM 2 only>>

#### Table 14.2-6.2.1 Raw cumulative incidence MMR during post-randomization Consolidation phase (ARM 2) - Subset of LSC sub-study Fulls Anslysis Set randomized to ARM 2

<< Programming note: Same shell as table 14.2-6.1, for LSC sub-study FAS ARM 2 only>>

<sup>-</sup> Confidence interval calculated as per Clopper-Pearson exact method.

#### Table 14.2-6.3 Raw cumulative incidence of MMR during re-treatment phase – Subset of Full Analysis Set entering the re-treatment phase

```
<<Programming note: Same shell as table 14.2-6.1, for re-treatment two arms >>
<<Programming note: From M27 onwards, arm2 patients should not be counted for the Total column>>
Use "Total*" for Total column and add footnote:
"* For month 27 onwards, only Arm1 patients considered for Total in percentages denominator."
```

#### Table 14.2-6.4 Raw cumulative incidence of MMR during re-treatment phase, SDV sensitivity – Subset of Full Analysis Set entering the re-treatment phase

```
<< Programming note: Same shell as Table 14.2-6.3, for SDV sensitivity analysis>>
Add footnote:
- SDV sensitivity: Excluding patient visits involved in SDV issues during final data review due to COVID-19.
```

# Table 14.2-7.1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase – Full Analysis Set

<< Programming note: Same shell as table 14.2-6.1, for MR4.0>>

#### Table 14.2-7.1.1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase – LSC sub-study Full Analysis Set

<< Programming note: Same shell as table 14.2-6.1.1, for MR 4.0>>

#### Table 14.2-7.2 Raw cumulative incidence of MR 4.0 during post-randomization consolidation phase (ARM 2) – Subset of Full Analysis Set randomized to ARM 2

< Programming note: < Same shell as table 14.2-6.2, for MR4.0 ARM 2 only>>

#### Table 14.2-7.2.1 Raw cumulative incidence of MR 4.0 during post-randomization consolidation phase (ARM 2) – Subset of LSC sub-study Full Analysis Set randomized to ARM 2

<< Programming note: Same shell as table 14.2-6.2.1, for MR4.0>>

### Table 14.2-7.3 Raw cumulative incidence of MR 4.0 during re-treatment phase – Subset of Full Analysis Set entering the re-treatment phase

```
<<Pre>rogramming note: Same shell as table 14.2-6.3, for MR 4.0 two arms >>
<<Pre><<Pre>counted for the Total column>>
Use "Total*" for Total column and add footnote:
"* For month 27 onwards, only Arm1 patients considered for Total in percentages denominator."
```

### Table 14.2-7.4 Raw cumulative incidence of MR 4.0 during re-treatment phase, SDV sensitivity – Subset of Full Analysis Set entering the re-treatment phase

```
<< Programming note: Same shell as Table 14.2-7.3, for SDV sensitivity analysis>>
Add footnote:
- SDV sensitivity: Excluding patient visits involved in SDV issues during final data review due to COVID-19.
```

# Table 14.2-8.1 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase – Full Analysis Set

<< Programming note: Same shell as table 14.2-6.1, for MR4.5 >>

# Table 14.2-8.1.1 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase – LSC sub-study Full Analysis Set

<< Programming note: Same shell as table 14.2-6.1, for MR 4.5>>

Table 14.2-8.2 Raw cumulative incidence of MR 4.5 during post-randomization consolidation phase (ARM 2) - Subset of Full Analysis Set randomized to Arm 2

<< Programming note: Same shell as table 14.2-6.2, for MR4.5 ARM 2 >>

Table 14.2-8.2.1 Raw cumulative incidence of MR 4.5 during post-randomization consolidation phase (ARM 2)
- Subset of LSC sub-study Full Analysis Set randomized to Arm 2

<< Programming note: Same shell as table 14.2-6.2.1, for MR 4.5 ARM 2>>

#### Table 14.2-8.3 Raw cumulative incidence of MR 4.5 during re-treatment phase - Subset of Full Analysis Set entering the re-treatment phase

```
<<Pre>rogramming note: Same shell as table 14.2-6.3, for MR 4.5 two arms >>
<<Pre><<Pre>counted for the Total column>>
Use "Total*" for Total column and add footnote:
"* For month 27 onwards, only Arm1 patients considered for Total in percentages denominator."
```

### Table 14.2-8.4 Raw cumulative incidence of MR 4.5 during re-treatment phase, SDV sensitivity - Subset of Full Analysis Set entering the re-treatment phase

<< Programming note: Same shell as Table 14.2-8.3, for SDV sensitivity analysis>>
Add footnote:

#### By halving time of BCR-ABL (IS) ratio

#### Table 14.2-9.1 Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase by halving time of BCR-ABL (IS) ratio – Full Analysis Set

| <pre>Halving time &lt;= 3 months / Halving time &gt; 3 months</pre> | Arm 1<br>N=xx | Arm 2<br>N=xx | Randomized<br>N=xx | Not Randomized N=xx | All patients<br>N=xx |
|---|---|---|---|---|---|
| Major molecular response at baseline | | | | | |
| Number of responders | xx | XX | XX | XX | XX |
| Percentage (95% CI) | xx (xx.x, xx.x) | xx (xx.x, xx.x) | xx (xx.x, xx.x) | xx (xx.x, xx.x) | xx (xx.x, xx.x) |
| Cumulative major molecular response up to 3 months (Day 91) | | | | | |
| Cumulative number of responders | XX | XX | XX | XX | XX |
| Cumulative percentage (95% CI) | xx (xx.x, xx.x) | xx ( $xx.x$ , $xx.x$ ) | xx (xx.x, xx.x) | xx ( $xx.x$ , $xx.x$ ) | xx (xx.x, xx.x) |
| Repeat for all time-points | | | | | |
| ••• | | | | | |
| Cumulative major molecular response up to 24 months (Day 730) | | | | | |
| Cumulative number of responders | XX | XX | XX | XX | XX |
| Cumulative percentage (95% CI) | xx (xx.x, xx.x) | xx (xx.x, xx.x) | xx (xx.x, xx.x) | xx (xx.x, xx.x) | xx (xx.x, xx.x) |

<sup>-</sup> Percentage based on the number of patients included in the analysis population (N)

#### << Programming note:

#### Table 14.2-9.1.1 Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase by halving time of BCR-ABL (IS) ratio – LSC sub-study Full Analysis Set

<< Programming note: Same shell as table 14.2-9.1, for LSC sub-study FAS>>

<sup>-</sup> Confidence Interval calculated as per Clopper-Pearson exact method

<sup>-</sup>Refer to the programming note of table 14.2-6.1.>>

Table 14.2-9.2 Raw cumulative incidence of MMR during post-randomization consolidation phase (ARM 2) by halving time of BCR-ABL (IS) ratio - Subset of Full Analysis Set randomized to Arm 2

| Arm 2<br>N=xx |
|-----------------------|
| XX |
| xx (xx.x, xx.x) |
| xx<br>xx (xx.x, xx.x) |
| WW |
| xx<br>xx (xx.x, xx.x) |

<sup>-</sup> Percentage based on the number of patients included in the analysis population (N)

<sup>-</sup> Confidence Interval calculated as per Clopper-Pearson exact method

# Table 14.2-9.2.1 Raw cumulative incidence of MMR during post-randomization consolidation phase (ARM 2) by halving time of BCR-ABL (IS) ratio - Subset of LSC sub-study Full Analysis Set randomized to Arm 2

<< Programming note: Same shell as table 14.2-9.2, for LSC sub-study FAS>>

#### Table 14.2-9.3 Raw cumulative incidence of MMR during re-treatment phase by halving time of BCR-ABL (IS) ratio – Subset of Full Analysis Set entering the re-treatment phase

<< Programming note: Same shell as table 14.2-9.1, for Re-treatment two arms >>
<<Programming note: From M27 onwards, arm2 patients should not be counted for the Total column>>
Use "Total\*" for Total column and add footnote:
"\* For month 27 onwards, only Arm1 patients considered for Total in percentages denominator."

Table 14.2-10.1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase by halving time of BCR-ABL (IS) ratio – Full Analysis Set

<< Programming note: Same shell as table 14.2-9.1, for MR 4.0 >>

Table 14.2-.10.1.1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase by halving time of BCR-ABL (IS) ratio – LSC sub-study Full Analysis Set

<< Programming note: Same shell as table 14.2-9.1.1, for MR 4.0 >>

Table 14.2-10.2 Raw cumulative incidence of MR 4.0 during post-randomization consolidation phase (ARM 2) by halving time of BCR-ABL (IS) ratio - Subset of Full Analysis Set randomized to Arm 2

<< Programming note: Same shell as table 14.2-9.2, for MR 4.0 ARM 2>>

Table 14.2-10.2.1 Raw cumulative incidence of MR 4.0 during post-randomization consolidation phase (ARM 2) by halving time of BCR-ABL (IS) ratio - Subset of LSC sub-study Full Analysis Set randomized to Arm 2

<< Programming note: Same shell as table 14.2-9.2.1, for MR 4.0 ARM 2>>

Table 14.2-10.3 Raw cumulative incidence of MR4.0 during re-treatment phase by halving time of BCR-ABL (IS) ratio – Subset of Full Analysis Set entering the re-treatment phase

<< Programming note: Same shell as table 14.2-9.3, for MR4.0 two arms >>
<<Programming note: From M27 onwards, arm2 patients should not be counted for the Total column>>
Use "Total\*" for Total column and add footnote:

"\* For month 27 onwards, only Arm1 patients considered for Total in percentages denominator."

#### Table 14.2-11.1 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase by halving time of BCR-ABL (IS) ratio – Full Analysis Set

<< Programming note: Same shell as table 14.2-9.1, for MR 4.5 >>

Table 14.2-.11.1.1 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase by halving time of BCR-ABL (IS) ratio – LSC sub-study Full Analysis Set

<< Programming note: Same shell as table 14.2-9.1.1, for MR 4.5 >>

Table 14.2-11.2 Raw cumulative incidence of MR 4.5 during post-randomization consolidation phase (ARM 2) by halving time of BCR-ABL (IS) ratio - Subset of Full Analysis Set randomized to Arm 2

<< Programming note: Same shell as table 14.2-9.2, for MR 4.5 ARM 2>>

Table14.2-11.2.1 Raw cumulative incidence of MR 4.5 during post-randomization consolidation phase (ARM 2) by halving time of BCR-ABL (IS) ratio - Subset of LSC sub-study Full Analysis Set randomized to Arm 2

<< Programming note: Same shell as table 14.2-9.2.1, for MR 4.5 ARM 2>>

Table 14.2-11.3 Raw cumulative incidence of MR4.5 during re-treatment phase by halving time of BCR-ABL (IS) ratio – Subset of Full Analysis Set entering the re-treatment phase

<< Programming note: Same shell as table 14.2-9.3, for MR4.5 two arms >>
<<Pre><<Pre><<Pre>counted for the Total column>>

```
{\it Use} "Total*" for Total column and add footnote:
```

"\* For month 27 onwards, only Arm1 patients considered for Total in percentages denominator."

#### By BCR-ABL (IS) ratio at Month 3

# Table 14.2-12.1 Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase by BCR-ABL (IS) ratio at Month 3 – Full Analysis Set

<< Programming note:

```
<< Same shell as table 14.2-9.1, with the following subgroups: BCR-ABL (IS) at Month 3 <= 0.005 BCR-ABL (IS) at Month 3 > 0.005>>
```

### Table 14.2-12.1.1 Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase by BCR-ABL (IS) ratio at Month 3 – LSC sub-study Full Analysis Set

<< Programming note:

```
<< Same shell as table 14.2-9.1.1, with the following subgroups: BCR-ABL (IS) at Month 3 <= 0.005 BCR-ABL (IS) at Month 3 > 0.005>>
```

# Table 14.2-12.2 Raw cumulative incidence of MMR during post-randomization consolidation phase (ARM 2) by BCR-ABL (IS) ratio at Month 3 - Subset of Full Analysis Set randomized to Arm 2

```
<< Programming note: Same shell as table 14.2-9.2, with the following subgroups: BCR-ABL (IS) at Month 3 <= 0.005 BCR-ABL (IS) at Month 3 > 0.005>>
```

### Table 14.2-12.2.1 Raw cumulative incidence of MMR during post-randomization consolidation phase (ARM 2) by BCR-ABL (IS) ratio at Month 3 - Subset of LSC sub-study Full Analysis Set randomized to Arm 2

```
<< Programming note: Same shell as table 14.2-9.2.1, with the following subgroups: BCR-ABL (IS) at Month 3 <= 0.005 BCR-ABL (IS) at Month 3 > 0.005>>
```

# Table 14.2-12.3 Raw cumulative incidence of MMR during re-treatment phase by BCR-ABL (IS) ratio at Month 3 – Subset of Full Analysis Set entering the re-treatment phase

```
<< Programming note: Same shell as table 14.2-9.2.3,
with the following subgroups:
BCR-ABL (IS) at Month 3 <= 0.005
BCR-ABL (IS) at Month 3 > 0.005>>

<<Pre><<Pre>C<Programming note: From M27 onwards, arm2 patients should not be counted for the Total column>>
Use "Total*" for Total column and add footnote:
"* For month 27 onwards, only Arm1 patients considered for Total in percentages denominator."
```

Table 14.2-13.1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase by BCR-ABL (IS) ratio at Month 3 – Full Analysis Set

<< Programming note: Same shell as table 14.2-12.1, for MR4.0 >>

Table 14.2-13.1.1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase by BCR-ABL (IS) ratio at Month 3 – LSC sub-study Full Analysis Set

<< Programming note: Same shell as table 14.2-12.1.1, for MR4.0 >>

Table 14.2-13.2 Raw cumulative incidence of MR 4.0 during post-randomization consolidation phase (ARM 2) by BCR-ABL (IS) ratio at Month 3 - Subset of Full Analysis Set randomized to Arm 2

<< Programming note: Same shell as table 14.2-12.2, for MR4.0 >>

Table 14.2-13.2.1 Raw cumulative incidence of MR 4.0 during post-randomization consolidation phase (ARM 2) by BCR-ABL (IS) ratio at Month 3 - Subset of LSC sub-study Full Analysis Set randomized to Arm 2

<< Programming note: Same shell as table 14.2-12.2.1, for MR4.0 >>

Table 14.2-13.3 Raw cumulative incidence of MR 4.0 during re-treatment phase by BCR-ABL (IS) ratio at Month 3 – Subset of Full Analysis Set entering the re-treatment phase

<<Pre><< Programming note: Same shell as table 14.2-12.3, for MR4.0 >>
<<Pre><<Pre><<Pre>Counted for the Total column column and add footnote:
"\* For month 27 onwards, only Arm1 patients considered for Total in percentages denominator."

Table 14.2-14.1 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase by BCR-ABL (IS) ratio at Month 3 – Full Analysis Set

<< Programming note: Same shell as table 14.2-12.1, for MR4.5 >>

Table 14.2-14.1.1 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase by BCR-ABL (IS) ratio at Month 3 – LSC sub-study Full Analysis Set

<< Programming note: Same shell as table 14.2-12.1.1, for MR4.5 >>

Table 14.2-14.2 Raw cumulative incidence of MR 4.5 during post-randomization consolidation phase (ARM 2) by BCR-ABL (IS) ratio at Month 3 - Subset of Full Analysis Set randomized to Arm 2

Programming note:

Table 14.2-14.2.1 Raw cumulative incidence of MR 4.5 during post-randomization consolidation phase (ARM 2) by BCR-ABL (IS) ratio at Month 3 - Subset of LSC sub-study Full Analysis Set randomized to Arm 2

<< Programming note: Same shell as table 14.2-12.2.1, for MR4.5 >>

Table 14.2-14.3 Raw cumulative incidence of MR 4.5 during re-treatment phase by BCR-ABL (IS) ratio at Month 3 – Subset of Full Analysis Set entering the re-treatment phase

<< Programming note: Same shell as table 14.2-12.3, for MR4.5 >>
<<Programming note: From M27 onwards, arm2 patients should not be counted for the Total column>>
Use "Total\*" for Total column and add footnote:
"\* For month 27 onwards, only Arm1 patients considered for Total in percentages denominator."

#### By Sokal Risk category

### Table 14.2-15.1 Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase by Sokal Risk category– Full Analysis Set

| Low risk (<0.8) Inermediate risk (>=0.8 - <=1.2) High risk (>1.2) | Arm 1<br>N=xx | Arm 2<br>N=xx | Randomized<br>N=xx | Not Randomized N=xx | All patients<br>N=xx |
|---|---|---|---|---|---|
| Major molecular response at baseline<br>Number of responders<br>Percentage (95% CI) | xx<br>xx (xx.x, xx.x) | xx<br>xx (xx.x, xx.x) | xx<br>xx (xx.x, xx.x) | xx<br>xx (xx.x, xx.x) | xx<br>xx (xx.x, xx.x) |
| Cumulative major molecular response up to 3 months (Day 91) Cumulative number of responders Cumulative percentage (95% CI) | xx<br>xx (xx.x, xx.x) | xx<br>xx (xx.x, xx.x) | xx<br>xx (xx.x, xx.x) | xx<br>xx (xx.x, xx.x) | xx<br>xx (xx.x, xx.x) |
| Repeat for all time-points | | | | | |
| Cumulative major molecular response up to 24 months (Day 730) Cumulative number of responders Cumulative percentage (95% CI) | xx<br>xx (xx.x, xx.x) | xx<br>xx (xx.x, xx.x) | xx<br>xx (xx.x, xx.x) | xx<br>xx (xx.x, xx.x) | xx<br>xx (xx.x, xx.x) |

<sup>-</sup> Percentage based on the number of patients included in the analysis population (N)

#### Table 14.2-15.2 Raw cumulative incidence of MR4.0 during pre-randomization Induction/Consolidation phase by Sokal Risk category– Full Analysis Set

<< Programming note: Same shell as table 14.2-15.1, for MR4.0>>

<sup>-</sup> Confidence Interval calculated as per Clopper-Pearson exact method

# Table 14.2-15.3 Raw cumulative incidence of MR4.5 during pre-randomization Induction/Consolidation phase by Sokal Risk category– Full Analysis Set

<< Programming note: Same shell as table 14.2-15.1, for MR4.5>>

#### By Time since initial diagnosis of CML

### Table 14.2-16.1 Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase by time since initial diagnosis of CML- Full Analysis Set

| <pre>&lt;2 years 2 to 4 years 4 to 6 years 6 to 8 years</pre> | | | | | |
|---|---|---|---|---|---|
| 8 to 10 years | | _ | | | |
| 10 to 12 years | Arm 1 | Arm 2 | Randomized | Not Randomized | All patients |
| >= 12 years | N=xx | N=xx | N=xx | N=xx | N=xx |
| Major molecular response at baseline | | | | | |
| Number of responders | XX | XX | XX | XX | XX |
| Percentage (95% CI) | xx (xx.x, xx.x) | xx (xx.x, xx.x) | xx (xx.x, xx.x) | xx (xx.x, xx.x) | xx (xx.x, xx.x) |
| Cumulative major molecular response up to 3 months (Day 91) Cumulative number of responders Cumulative percentage (95% CI) | xx<br>xx (xx.x, xx.x) | xx<br>xx (xx.x, xx.x) | xx<br>xx (xx.x, xx.x) | xx<br>xx (xx.x, xx.x) | xx<br>xx (xx.x, xx.x) |
| Repeat for all time-points | | | | | |
| Cumulative major molecular response up to 24 months (Day 730) Cumulative number of responders | xx | xx | xx | xx | xx |
| Cumulative percentage (95% CI) | xx (xx.x, xx.x) | xx (xx.x, xx.x) | xx (xx.x, xx.x) | xx (xx.x, xx.x) | xx (xx.x, xx.x) |

<sup>-</sup> Percentage based on the number of patients included in the analysis population (N)

<sup>-</sup> Confidence Interval calculated as per Clopper-Pearson exact method.

Table 14.2-16.2 Raw cumulative incidence of MR4.0 during pre-randomization Induction/Consolidation phase by time since initial diagnosis of CML – Full Analysis Set

<< Programming note: Same shell as table 14.2-16.1, for MR4.0>>

Table 14.2-16.3 Raw cumulative incidence of MR4.5 during pre-randomization Induction/Consolidation phase by time since initial diagnosis of CML – Full Analysis Set

<< Programming note: Same shell as table 14.2-16.1, for MR4.5>>
#### **Suboptimal response**

Table 14.2-17.1 Suboptimal response up to 24 months of pre-randomization Induction/Consolidation phase - Full Analysis Set patients who prematurely discontinued the pre-randomization Induction/Consolidation phase

| Criteria | Arm 1<br>N=xx | Arm 2<br>N=xx | Randomized<br>N=xx | Not Randomized<br>N=xx | Total<br>N=xx |
|---|---|---|---|---|---|
| At least one criterion of suboptimal response n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| loss of CHR - n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| loss of CCyR - n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| loss of MMR - n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| no MMR up to Month 24 - n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

<sup>-</sup> Percentage based on the number of patients included in the analysis population (N).

- Patient # randomized to Arm 1 at and discontinued Ind/cons at the same day for

#### << Programming note:

- The loss of CHR, CCyR and MMR should be displayed only if they occurred before or at Month 24 (ie 730 days).
- no MMR up to Month 24 means no MMR up to 730 days.>>

<sup>-</sup> CHR: Complete hematologic response = normalization of hematopoiesis.

<sup>-</sup> CCyR: Complete cytogenetic response.

# Table 14.2-17.2 Suboptimal response up to 12 months of post-randomization Consolidation phase (ARM 2) - Subset of Full Analysis Set patients who prematurely discontinued the Induction/Consolidation phase randomized to Arm 2

| Criteria | N=XX |
|-----------------------------------------------------|-----------|
| At least one criterion of suboptimal response n (%) | xx (xx.x) |
| loss of CHR - n (%) | xx (xx.x) |
| loss of CCyR - n (%) | xx (xx.x) |
| loss of MMR - n (%) | xx (xx.x) |
| no MMR up to Month 12* - n (%) | xx (xx.x) |

<sup>-</sup> Percentage based on the number of patients included in the analysis population (N).

#### << Programming note:

### Table 14.2-18.1 Suboptimal response up to 24 months of pre-randomization Induction/Consolidation phase - Full Analysis Set

<< Programming note:

- Same as Table 14.2-17.1 on all treated patients.>>

### Table 14.2-18.2 Suboptimal response up to 12 months of post-randomization Consolidation phase - Subset of Full Analysis Set, randomized to ARM 2

<< Programming note:

- Same as Table 14.2-17.2 on all treated patients.>>

<sup>-</sup> CHR: Complete hematologic response = normalization of hematopoiesis.

<sup>-</sup> CCyR: Complete cytogenetic response.

<sup>\*</sup> After Randomization.

<sup>- 15</sup> patients from ARM 2 discontinued during post-Randomization Consolidation phase.

<sup>-</sup> The loss of CHR, CCyR and MMR should be displayed only if they occurred before or at Month 12 (ie 365 days) 12 months after randomization.

<sup>-</sup> no MMR up to Month 12 means no MMR up to 365 days (12 months after randomization).

#### **Kinetics**

Table 14.2-19.1 Kinetics of BCR-ABL (IS) ratio during pre-randomization Induction/Consolidation phase – Full Analysis Set

| | Arm 1<br>N=xx | Arm 2<br>N=xx | Randomized<br>N=xx | Not Randomized N=xx | Total<br>N=xx |
|---|---|---|---|---|---|
| BCR-ABL (IS) (%) at Baseline | | | | | |
| n | xx | xx | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | X.XX | X.XX | X.XX | X.XX | X.XX |
| 25th Percentile | XX.X | XX.X | XX.X | XX.X | XX.X |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| 75th Percentile | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min-Max | xx.x-xx.x | xx.x-xx.x | xx.x-xx.x | xx.x-xx.x | xx.x-xx.x |
| BCR-ABL (IS) (%) at Month 3 | | | | | |
| n | XX | XX | XX | XX | XX |
| •• | | | | | |
| Min-Max | xx.x-xx.x | xx.x-xx.x | xx.x-xx.x | XX.X-XX.X | xx.x-xx.x |
| Repeat at each time-point | | | | | |
| BCR-ABL (IS) (%) at Month 36 | | | | | |
| n | XX | XX | XX | XX | XX |
| 75th Percentile<br>Min-Max | xx.x<br>xx.x-xx.x | xx.x<br>xx.x-xx.x | xx.x<br>xx.x-xx.x | xx.x<br>xx.x-xx.x | xx.x<br>xx.x-xx.x |

<sup>-</sup> The last value of BCR-ABL (IS) ratio per time-window is displayed in this table.

Table 14.2-19.1.1 Kinetics of BCR-ABL (IS) ratio during pre-randomization Induction/Consolidation phase – LSC sub-study Full Analysis Set

<< Programming note: Same shell as table 14.2-19.1, for LSC sub-study FAS>>

Table 14.2-19.2 Kinetics of BCR-ABL (IS) ratio during post-randomization consolidation phase (ARM 2) – Subset of Full Analysis Set randomized to Arm 2

| | | | | | | N=xx |
|----------|-------|-----|----|-------|----|----------------|
| BCR-ABL | (IS) | (%) | at | Month | 27 | |
| n | | | | | | XX |
| Mean | | | | | | XX.X |
| SD | | | | | | X.XX |
| 25th Per | centi | lle | | | | XX.X |
| Median | | | | | | XX.X |
| 75th Per | centi | lle | | | | XX.X |
| Min Max | | | | | | xx.x -xx.x |
| BCR-ABL | (IS) | (응) | at | Month | 30 | xx |
| Min Max | | | | | | <br>xx.x -xx.x |
| BCR-ABL | (IS) | (%) | at | Month | 33 | |
| n | | | | | | XX |
| • • • | | | | | | • • • |
| BCR-ABL | (IS) | (%) | at | Month | 36 | |
| n | | | | | | XX |
| Min Max | | | | | | xx.x -xx.x |

<sup>-</sup> The last value of BCR-ABL (IS) ratio per time-window is displayed in this table.

## Table 14.2-19.2.1 Kinetics of BCR-ABL (IS) ratio during post-randomization consolidation phase (ARM 2) – Subset of LSC sub-study Full Analysis Set randomized to Arm 2

<< Programming note: Same shell as table 14.2-19.2, for LSC sub-study FAS>>

Table 14.2-19.3 Kinetics of BCR-ABL (IS) ratio during TFR phase – Subset of Full Analysis Set entering the TFR phase

| · | Arm 1 | Arm 2 | Total |
|------------------------------------------|-----------|-----------|-----------|
| | N=xx | N=xx | N=xx |
| BCR-ABL (IS) (%) at Month 1 | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | X.XX | X.XX | X.XX |
| 25th Percentile | XX.X | XX.X | XX.X |
| Median | XX.X | XX.X | XX.X |
| 75th Percentile | XX.X | XX.X | XX.X |
| Min-Max | xx.x-xx.x | xx.x-xx.x | xx.x-xx.x |
| Repeat at each time-point every 1 month | | | |
| BCR-ABL (IS) (%) at Month 6 | | | |
| n | XX | XX | XX |
| ••• | ••• | • • • | ••• |
| Min-Max | xx.x-xx.x | xx.x-xx.x | xx.x-xx.x |
| Repeat at each time-point every 2 months | | | |
| BCR-ABL (IS) (%) at Month 12 | | | |
| n | XX | Xx | XX |
| ••• | • • • | | |
| Min-Max | xx.x-xx.x | xx.x-xx.x | xx.x-xx.x |

| Novartis | Confidential<br>6-May-2021 (14:35) | | Protocol No CAMN107AICO |
|---|---|---|---|
| RAP Module 7.1 | 0-May-2021 (14.33) | | Protocol No CAMN107AIC0 |
| Repeat at each time-point every 3 months | | | |
| BCR-ABL (IS) (%) at Month 24 | | | |
| n | XX | Xx | XX |
| ••• | • • • | • • • | • • • |
| Min-Max | xx.x-xx.x | xx.x-xx.x | xx.x-xx.x |
| Repeat at each time-point every 3 months | | | |
| BCR-ABL (IS) (%) at Month 36 | | | |
| n | XX | | XX |
| ••• | • • • | | • • • |
| Min-Max | xx.x-xx.x | | xx.x-xx.x |

<sup>-</sup> Patients randomized to Arm 2 have a maximum of 24 months of TFR phase.

<sup>-</sup> The last value of BCR-ABL (IS) ratio per time-window is displayed in this table.

Table 14.2-19.4 Kinetics of BCR-ABL (IS) ratio during re-treatment phase – Subset of Full Analysis Set entering the re-treatment phase

| · | Arm 1 | Arm 2 | Total |
|------------------------------------------|-----------|-----------|-----------|
| | N=xx | N=xx | N=XX |
| BCR-ABL (IS) (%) at Day 1 | | | |
| n | XX | Xx | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | X.XX | X.XX | X.XX |
| 25th Percentile | XX.X | XX.X | XX.X |
| Median | xx.x | XX.X | XX.X |
| 75th Percentile | xx.x | xx.x | XX.X |
| Min-Max | xx.x-xx.x | xx.x-xx.x | xx.x-xx.x |
| BCR-ABL (IS) (%) at Week 6 | | | |
| n | xx | Xx | xx |
| ••• | | | |
| Min-Max | xx.x-xx.x | xx.x-xx.x | xx.x-xx.x |
| BCR-ABL (IS) (%) at Month 3 | | | |
| n | xx | Xx | XX |
| ••• | • • • | | ••• |
| Min-Max | xx.x-xx.x | xx.x-xx.x | xx.x-xx.x |
| Repeat at each time-point every 3 months | | | |
| BCR-ABL (IS) (%) at Month 36 | | | |
| n | XX | | xx |
| ••• | | | ••• |
| Min-Max | xx.x-xx.x | | xx.x-xx.x |

<sup>-</sup> Patients randomized to Arm 2 have a maximum of 24 months of re-treatment phase.

<sup>-</sup> The last value of BCR-ABL (IS) ratio per time-window is displayed in this table

## Table 14.2-19.5 Kinetics of BCR-ABL (IS) ratio during TFR phase, SDV sensitivity — Subset of Full Analysis Set entering the TFR phase

<< Programming note: Same shell as Table 14.2-19.3, for SDV sensitivity analysis>> Add footnote:

- SDV sensitivity: Excluding patient visits involved in SDV issues during final data review due to COVID-19.

### Table 14.2-19.6 Kinetics of BCR-ABL (IS) ratio during re-treatment phase, SDV sensitivity - Subset of Full Analysis Set entering the re-treatment phase

<< Programming note Same shell as Table 14.2-19.4, for SDV sensitivity analysis>> Add footnote:

- SDV sensitivity: Excluding patient visits involved in SDV issues during final data review due to COVID-19.

#### Patients Not reaching MMR/ MR 4.0 / MR 4.5

### Table 14.2-20.1 Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase - Full Analysis Set patients not reaching MMR at baseline

<< Programming note:

-Same shell as cumulative incidence of MMR table (14.2-6.1) but performed on the subset of subjects not reaching MMR at baseline (i.e. time-to-first MMR not equal to 0).
-Remove "Major molecular response at baseline".

### Table 14.2-20.2 Raw cumulative incidence of MMR during post-randomization Consolidation phase (ARM 2) - Subset of Full Analysis Set patients not reaching MMR at baseline, randomized to ARM 2

<< Programming note:

-Same shell as cumulative incidence of MMR table (table 14.2-6.2) but performed on the subset of subjects not reaching MMR at baseline (i.e. time-to-first MMR not equal to 0).

### Table 14.2-21.1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase - Full Analysis Set patients not reaching MR 4.0 at baseline

<< Programming note:

-Same shell as cumulative incidence of MR 4.0 table (14.2-7.1) but performed on the subset of subjects not reaching 4.0 at baseline (i.e. time-to-first MR 4.0 not equal to 0).
-Remove "Molecular response 4.0 at baseline". >>

### Table 14.2-21.2 Raw cumulative incidence of MR 4.0 during post-randomization Consolidation phase (ARM 2) - Subset of Full Analysis Set patients not reaching MR 4.0 at baseline, randomized to ARM 2

<< Programming note:

-Same shell as cumulative incidence of MR 4.0 table (table 14.2-8.2) but performed on the subset of subjects not reaching MR 4.0 at baseline (i.e. time-to-first MR 4.0 not equal to 0).

### Table 14.2-22.1 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase - Full Analysis Set patients not reaching MR 4.5 at baseline

<< Programming note:

-Same shell as cumulative incidence of MR 4.5 table (table 14.2-9.1) but performed on the subset of subjects not reaching MR 4.5 at baseline (i.e. time-to-first MR 4.5 not equal to 0).

-Remove "Molecular response 4.5 at baseline". >>

### Table 14.2-22.2 Raw cumulative incidence of MR 4.5 during post-randomization Consolidation phase (ARM 2) - Subset of Full Analysis Set patients not reaching MR 4.5 at baseline, randomized to ARM 2

<< Programming note:

-Same shell as cumulative incidence of MR 4.5 table (table 14.2-9.2) but performed on the subset of subjects not reaching MR 4.5 at baseline (i.e. time-to-first MR 4.5 not equal to 0).

-Refer to the programming note of table 14.2-6.2.>>

### Table 14.2-22.3 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase

- Full Analysis Set patients not reaching MMR at baseline

<<pre><<Pre>rogramming note:

-Same shell as cumulative incidence of MR 4.0 table (table 14.2-7.1) but performed on the subset of subjects not reaching MMR at baseline.>>

### Table 14.2-22.4 Raw cumulative incidence of MR 4.0 during post-randomization Consolidation phase (ARM 2)

- Subset of Full Analysis Set patients not reaching MMR at baseline, randomized to ARM 2

<< Programming note:

-Same shell as cumulative incidence of MR 4.0 table (table 14.2-7.2) but performed on the subset of subjects not reaching MMR at baseline.>>

### Table 14.2-22.5 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase - Full Analysis Set patients not reaching MMR at baseline

<< Programming note:

-Same shell as cumulative incidence of MR 4.5 table (table 14.2-8.1) but performed on the subset of subjects not reaching MMR at baseline.>>

### Table 14.2-22.6 Raw cumulative incidence of MR 4.5 during post-randomization Consolidation phase (ARM 2) - Subset of Full Analysis Set patients not reaching MMR at baseline, randomized to ARM 2

<< Programming note:

-Same shell as cumulative incidence of MR 4.5 table (table 14.2-8.2) but performed on the subset of subjects not reaching MMR at baseline.>>

#### By BCR-ABL(IS) ratio at baseline

### Table 14.2-23.1 Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase by BCR-ABL(IS) ratio at baseline - Full Analysis Set

| BCR-ABL(IS) ratio >0.1% - ≤1% / BCR-ABL(IS) ratio >0.01% -≤0.1% | Arm 1<br>N=xx | Arm 2<br>N=xx | Randomized<br>N=xx | Not Randomized<br>N=xx | Total<br>N=xx |
|---|---|---|---|---|---|
| Molecular response 4.0 at baseline | | | | | |
| Number of responders | XX | XX | XX | XX | XX |
| Percentage (95% CI) | xx (xx.x, xx.x) | xx (xx.x, xx.x) | xx (xx.x, xx.x) | xx (xx.x, xx.x) | xx (xx.x, xx.x) |
| Cumulative molecular response 4.0 up to 3 months (Day 91) Cumulative number of responders | xx | xx | xx | xx | xx |
| Cumulative percentage (95% CI) | xx (xx.x, xx.x) | xx (xx.x, xx.x) | xx (xx.x, xx.x) | xx (xx.x, xx.x) | xx (xx.x, xx.x) |
| Cumulative molecular response 4.0 up to 6 months (Day 182) | | | | | |
| ••• | • • • | • • • | • • • | • • • | • • • |
| Repeat until 24 months | | | | | |
| Cumulative molecular response 4.0 up to 24 months (Day 730) Cumulative number of responders | xx | xx | xx | xx | xx |
| Cumulative percentage (95% CI) | xx (xx.x, xx.x) | | | xx (xx.x, xx.x) | |

<sup>-</sup> Percentage based on the number of patients included in the analysis population (N)

#### << Programming note:

- Same shell as Table 4.8 but by BCR-ABL(IS) ratio (use MRCATBL = 2 for BCR-ABL(IS) ratio >0.1% -  $\leq$ 1%, and MRCATBL = 3 for BCR-ABL(IS) ratio >0.01% -  $\leq$ 0.1%)>

<sup>-</sup> Confidence Interval calculated as per Clopper-Pearson exact method

### Table 14.2-23.1.1 Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase by BCR-ABL (IS) ratio at baseline– LSC sub-study Full Analysis Set

<< Programming note: Same shell as table 14.2-23.1, for LSC sub-study FAS>>

### Table 14.2-23.2 Raw cumulative incidence of MMR during post-randomization consolidation phase (ARM 2) by BCR-BL(IS) ratio at baseline - Subset of Full Analysis Set, randomized to ARM 2

| BCR-ABL(IS) ratio >0.1% - ≤1% / BCR-ABL(IS) ratio >0.01% -≤0.1% | N=xx |
|---|---|
| Molecular response 4.0 at baseline | |
| Number of responders | XX |
| Percentage (95% CI) | xx (xx.x, xx.x) |
| Cumulative molecular response 4.0 up to 27 months (Day 822) Cumulative number of responders | xx |
| Cumulative percentage (95% CI) | xx (xx.x, xx.x) |
| Cumulative molecular response 4.0 up to 30 months (Day 913) | |
| Repeat until 36 months | |
| Cumulative molecular response 4.0 up to 36 months (Day 1096) | |
| Cumulative number of responders | XX |
| Cumulative percentage (95% CI) | xx (xx.x, xx.x) |

<sup>-</sup> Percentage based on the number of patients included in the analysis population (N)

#### << Programming note:

<sup>-</sup> Confidence Interval calculated as per Clopper-Pearson exact method

- Same shell as Table 4.8 but by BCR-ABL(IS) ratio (use MRCATBL = 2 for BCR-ABL(IS) ratio >0.1% -  $\leq$ 1%, and MRCATBL = 3 for BCR-ABL(IS) ratio >0.01% -  $\leq$ 0.1%)>>

Table 14.2-23.2.1 Raw cumulative incidence of MMR during post-randomization consolidation phase (ARM 2) by BCR-BL(IS) ratio at baseline - Subset of LSC sub-study Full Analysis Set, randomized to ARM 2

<< Programming note: Same shell as table 14.2-23.2, for LSC sub-study FAS ARM 2>>

Table 14.2-23.3 Raw cumulative incidence of MMR during re-treatment phase by BCR-BL(IS) ratio at baseline – Subset of Full Analysis Set entering the re-treatment phase

<< Programming note:

- Same shell as Table 14.2-23.1, but for re-treatment two arms >> Add footnote: \*For month 27 onwards, only Arm1 patients considered for Total in percentages denominator." Programing note added."

Table 14.2-24.1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase by BCR-ABL(IS) ratio at baseline - Full Analysis Set

<< Programming note: Same shell as table 14.2-23.1, for MR 4.0 >>

Table 14.2-24.1.1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase by BCR-ABL (IS) ratio at baseline– LSC sub-study Full Analysis Set

<< Programming note: Same shell as table 14.2-23.1.1, for MR 4.0 >>

Table 14.2-24.2 Raw cumulative incidence of MR 4.0 during post-randomization consolidation phase (ARM 2) by BCR-BL(IS) ratio at baseline - Subset of Full Analysis Set, randomized to ARM 2

<< Programming note: Same shell as table 14.2-24.2, for MR 4.0 >>

Table 14.2-24.2.1 Raw cumulative incidence of MR 4.0 during post-randomization consolidation phase (ARM 2) by BCR-BL(IS) ratio at baseline - Subset of LSC sub-study Full Analysis Set , randomized to ARM 2

<< Programming note: Same shell as table 14.2-24.2.1, for MR 4.0 >>

Table 14.2-24.3 Raw cumulative incidence of MR 4.0 during re-treatment phase by BCR-BL(IS) ratio at baseline – Subset of Full Analysis Set entering the re-treatment phase

<< Programming note: Same shell as table 14.2-24.3, for MR 4.0 >>
Add footnote: \*For month 27 onwards, only Arm1 patients considered for Total in percentages denominator." Programing note
added."

Table 14.2-25.1 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase by BCR-ABL(IS) ratio at baseline - Full Analysis Set

<< Programming note: Same shell as table 14.2-23.1, for MR 4.5 >>

Table 14.2-25.1.1 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase by BCR-ABL (IS) ratio at baseline– LSC sub-study Full Analysis Set

<< Programming note: Same shell as table 14.2-23.1.1, for MR 4.5 >>

Table 14.2-25.2 Raw cumulative incidence of MR 4.5 during post-randomization consolidation phase (ARM 2) by BCR-BL(IS) ratio at baseline - Subset of Full Analysis Set, randomized to ARM 2

<< Programming note: Same shell as table 14.2-24.2, for MR 4.5 >>

Table 14.2-25.2.1 Raw cumulative incidence of MR 4.5 during post-randomization consolidation phase (ARM 2) by BCR-BL(IS) ratio at baseline - Subset of LSC sub-study Full Analysis Set , randomized to ARM 2

<< Programming note: Same shell as table 14.2-24.2.1, for MR 4.5 >>

Table 14.2-25.3 Raw cumulative incidence of MR 4.5 during re-treatment phase by BCR-BL(IS) ratio at baseline – Subset of Full Analysis Set entering the re-treatment phase

<< Programming note: Same shell as table 14.2-24.3, for MR 4.5 >>
Add footnote: \*For month 27 onwards, only Arm1 patients considered for Total in percentages denominator." Programing note
added."

#### Loss of MMR/ MR 4.0, MR 4.5 during TFR

## Table 14.2-26.1 Raw cumulative loss of MMR during TFR phase –Subset of Full Analysis Set entering the TFR phase

| • | Arm 1<br>N=xx | Arm 2<br>N=xx | Total*<br>N=xx |
|---|---|---|---|
| Major molecular response at Baseline TFR | | | |
| Number of responders | XX | XX | XX |
| Percentage (95% CI) | xx ( $xx.x$ , $xx.x$ ) | xx (xx.x, xx.x) | xx (xx.x, xx.x) |
| Cumulative loss of major molecular response up to 1 month (Day 30) | | | |
| Cumulative number with loss | XX | XX | XX |
| Cumulative percentage (95% CI) | xx (xx.x, xx.x) | xx (xx.x, xx.x) | xx (xx.x, xx.x) |
| Repeat at each-time point every month | | | |
| Cumulative loss of major molecular response up to 6 months (Day 183) | | | |
| Cumulative number with loss | XX | XX | XX |
| Cumulative percentage (95% CI) | xx (xx.x, xx.x) | xx (xx.x, xx.x) | xx (xx.x, xx.x) |
| Repeat at each-time point every 2 months | | | |
| Cumulative loss of major molecular response up to 12 months (Day 365) | | | |
| Cumulative number with loss | xx | xx | XX |
| Cumulative percentage (95% CI) | xx ( $xx.x$ , $xx.x$ ) | xx (xx.x, xx.x) | xx (xx.x, xx.x) |
| Repeat at each-time point every 3 months | | | |
| Cumulative loss of major molecular response up to 36 months (Day 1096) | | | |
| Cumulative number with loss | XX | | XX |
| Cumulative percentage (95% CI) | xx (xx.x, xx.x) | | xx (xx.x, xx.x) |

<sup>-</sup> The baseline TFR corresponds to the last available assessment before or on the last day of study drug intake from induction/consolidation phase.

<sup>-</sup> Patients randomized to Arm 2 have a maximum of 24 months of TFR phase.

<sup>-</sup> Confidence interval calculated as per Clopper-Pearson exact method.

<sup>-</sup> Percentage based on the number of patients included in the analysis population (N).

<sup>\*</sup> For month 27 onwards, only Arm 1 patients considered for Total in percentages denominator.

#### << Programming note:

- -Cumulative number with response at Month x is obtained by counting all patients with a time to response in day before day x;
   Day x = round(30.4375\*months).
- -The percentage is obtained by dividing the number with response by N.>>

### Table 14.2-26.2 Raw cumulative loss of MR4.0 during TFR phase –Subset of Full Analysis Set entering the TFR phase

<< Programming note: Same shell as table 14.2-26.1 replacing "major molecular response" by "molecular response 4.0" >>
<<Programming note: From M27 onwards, Arm 2 patients should not be counted for the Total column>>

## Table 14.2-26.3 Raw cumulative loss of MR4.5 during TFR phase –Subset of Full Analysis Set entering the TFR phase with MR4.5

<< Programming note: Same shell as table 14.2-26.1 replacing "major molecular response" by "molecular response 4.5" >> << Programming note: From M27 onwards, Arm 2 patients should not be counted for the Total column>>

### Table 14.2-26.4 Raw cumulative loss of MMR during TFR phase, SDV sensitivity -Subset of Full Analysis Set entering the TFR phase

<< Programming note: Same shell as Table 14.2-26.1, for SDV sensitivity analysis>>
Add footnote:

- SDV sensitivity: Excluding patient visits involved in SDV issues during final data review due to COVID-19.

### Table 14.2-26.5 Raw cumulative loss of MR4.0 during TFR phase, SDV sensitivity –Subset of Full Analysis Set entering the TFR phase

<< Programming note: Same shell as Table 14.2-26.2, for SDV sensitivity analysis>> Add footnote:

- SDV sensitivity: Excluding patient visits involved in SDV issues during final data review due to COVID-19.

### Table 14.2-26.6 Raw cumulative loss of MR4.5 during TFR phase, SDV sensitivity –Subset of Full Analysis Set entering the TFR phase with MR4.5

<< Programming note: Same shell as Table 14.2-26.3, for SDV sensitivity analysis>> Add footnote:

- SDV sensitivity: Excluding patient visits involved in SDV issues during final data review due to COVID-19.

#### LSC substudy descriptives

Table 14.2-27.1 Descriptive Statistics for CD34 cells: Total percentage – LSC sub-study Full Analysis Set

| | Arm 1<br>N=xx | Arm 2<br>N=xx | Randomized<br>N=xx | Not<br>Randomized<br>N=xx | Total<br>N=xx |
|---|---|---|---|---|---|
| Baseline [1] | | | | | |
| n | xx | XX | XX | XX | XX |
| Mean | xx.x | XX.X | XX.X | XX.X | XX.X |
| SD | x.xx | X.XX | X.XX | X.XX | X.XX |
| Min | XX | XX | XX | XX | XX |
| 25th Percentile | XX.X | XX.X | XX.X | XX.X | XX.X |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| 75th Percentile | xx.x | XX.X | XX.X | XX.X | XX.X |
| Max | XX | XX | XX | XX | XX |
| Month 24 | | | | | |
| n | XX | XX | XX | XX | XX |
| • • • | • • • | | • • • | • • • | |
| Max | XX | XX | XX | XX | XX |
| Change from Baseline to Month 24 | | | | | |
| n | XX | XX | XX | XX | XX |
| ••• | • • • | • • • | • • • | • • • | • • • |
| Max | XX | XX | XX | XX | XX |
| Month 36 | | | | | |
| | • • • | • • • | • • • | • • • | • • • |
| Change from Baseline to Month 36 | | | | | |
| n | - | XX | XX | XX | XX |
| ••• | | | | | |
| Max | _ | XX | XX | XX | XX |

| Confidential<br>6-May-2021 (14:35) | | | Page 258<br>Protocol No CAMN107AIC0 | |
|---|---|---|---|---|
| VV | V V | VV | <b>V</b> V | xx |
| <br>xx | <br>XX | <br>XX | <br>XX | <br>xx |
| -<br> | xx<br> | xx<br><br>xx | xx<br><br>xx | xx<br><br>xx |
| | 6-May-2021 (14:35) | 6-May-2021 (14:35) | 6-May-2021 (14:35) | 6-May-2021 (14:35) |

<sup>[1]</sup> Baseline is defined as latest visit between Screening or Rescreening.

<sup>-</sup> Change from Baseline derived if both baseline and timepoint evaluation are available.

<sup>-</sup> Only available numeric values are presented.

Table 14.2-28.1 Descriptive Statistics for CD34+/CD38+ cells: Percentage from total CD34+ cells – LSC substudy Full Analysis Set

| - | Arm 1<br>N=xx | Arm 2<br>N=xx | Randomized<br>N=xx | Not<br>Randomized<br>N=xx | Total<br>N=xx | Comparison<br>p-value# |
|---|---|---|---|---|---|---|
| Baseline [1] | | | | | | |
| n | XX | XX | XX | XX | XX | |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | |
| SD | X.XX | X.XX | X.XX | X.XX | X.XX | |
| Min | XX | XX | XX | XX | XX | |
| 25th Percentile | XX.X | XX.X | XX.X | XX.X | XX.X | |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | |
| 75th Percentile | XX.X | XX.X | XX.X | XX.X | XX.X | |
| Max | XX | XX | XX | XX | XX | |
| Month 24 | | | | | | |
| n | XX | XX | XX | XX | XX | |
| ••• | | | | | | |
| Max | XX | XX | XX | XX | XX | |
| Change from Baseline to Month 24 | | | | | | |
| n | XX | XX | XX | XX | XX | 0.xxx |
| ••• | | | | | | 0.xxx |
| Max | XX | XX | XX | XX | XX | |
| Month 36 | | | | | | |
| | • • • | • • • | • • • | • • • | • • • | |
| Change from Baseline to Month 36 | | | | | | |
| n | - | XX | XX | | XX | |
| ••• | • • • | • • • | • • • | | • • • | |
| Max | _ | XX | XX | | XX | |
| EOP TFR | | | | | | |
| n | XX | XX | XX | | XX | |
| | • • • | • • • | • • • | | • • • | |
| Max | XX | XX | XX | | XX | |

|----------------|--------------------|-------------------------|
| RAP Module 7.1 | 6-May-2021 (14:35) | Protocol No CAMN107AIC0 |

| Change f | from Baseline to EOP T | 'FR | | | |
|----------|------------------------|-------|----|-------|-------|
| n | l | XX | XX | XX | XX |
| | • | • • • | | • • • | • • • |
| Ma | X | XX | XX | XX | XX |

<sup>[1]</sup> Baseline is defined as latest visit between Screening or Rescreening.

## Table 14.2-28.2 Descriptive Statistics for number of events sorted in CD34+/CD38+ cells – LSC sub-study Full Analysis Set

<< Programming note: Same shell as table 14.2-28.1 >>

<sup>-</sup> Change from Baseline derived if both baseline and timepoint evaluation are available.

<sup>-</sup> Only available numeric values are presented.

<sup>\$</sup> Comparison Rand. vs Not Rand. # P-value:independent t-test for means, Median test for medians.

<sup>\*</sup> p-value<0.05, \*\* p-value<0.01.

Table 14.2-28.3 Ph+ by HIS status, in CD34+/CD38+ cells - LSC sub-study Full Analysis Set

| • | Arm 1 | Arm 2 Random: | Randomized | mized Not Randomized | ized Total<br>N=xx |
|---|---|---|---|---|---|
| | N=xx | N=xx | N=xx | N=xx | |
| Baseline [1] | | | | | |
| Not Evaluable | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Negative | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Positive | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Missing | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Month 24 | | | | | |
| Not Evaluable | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Negative | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Positive | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Missing | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Month 36 | | | | | |
| Not Evaluable | _ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Negative | _ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Positive | _ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Missing | _ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| EOP TFR | | | | | |
| Not Evaluable | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Negative | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Positive | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Missing | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

<sup>[1]</sup> Baseline is defined as latest visit between Screening or Rescreening.

Table 14.2-28.4 Descriptive statistics of Ph+ in CD34+/CD38+ cells- LSC sub-study Full Analysis Set 
</ Programming note: Same shell as table 14.2-28.1 >>

Table 14.2-28.5 BCR-ABL by RT-PCR status, in CD34+/CD38+ cells – LSC sub-study Full Analysis Set 
</ Programming note: Same shell as table 14.2-28.3 >>

### Repeat for CD34+/CD38- cells:

Table 14.2-29.1 Descriptive Statistics for CD34+/CD38- cells: Percentage from total CD34+ cells – LSC substudy Full Analysis Set

<< Programming note: Same shell as table 14.2-28.1, exclude p-values >>

Table 14.2-29.2 Descriptive Statistics for number of events sorted in CD34+/CD38- cells – LSC sub-study Full Analysis Set

<< Programming note: Same shell as table 14.2-28.1, exclude p-values >>

Table 14.2-29.3 Ph+ by HIS status, in CD34+/CD38- cells – LSC sub-study Full Analysis Set 
</ Programming note: Same shell as table 14.2-28.3 >>

Table 14.2-29.5 BCR-ABL by RT-PCR status, in CD34+/CD38- cells – LSC sub-study Full Analysis Set 
</ Programming note: Same shell as table 14.2-28.3 >>

### Repeat for Immunophenotypically aberrant CD34+ cells:

Table 14.2-30.1 Descriptive Statistics for Immunophenotypically aberrant CD34+ cells: Percentage from total CD34+ cells –LSC sub-study Full Analysis Set

<< Programming note: Same shell as table 14.2-28.1, exclude p-values >>

Table 14.2-30.2 Descriptive Statistics for number of events sorted in Immunophenotypically aberrant CD34+ cells – LSC sub-study Full Analysis Set

<< Programming note: Same shell as table 14.2-28.1, exclude p-values >>

Table 14.2-30.3 Ph+ by HIS status, in Immunophenotypically aberrant CD34+ cells – LSC sub-study Full Analysis Set

<< Programming note: Same shell as table 14.2-28.3 >>

Table 14.2-30.4 Descriptive statistics of Ph+ in Immunophenotypically aberrant CD34+ cells– LSC sub-study Full Analysis Set

<< Programming note: Same shell as table 14.2-28.1 >>

Table 14.2-30.5 BCR-ABL by RT-PCR status, in Immunophenotypically aberrant CD34+ cells – LSC sub-study Full Analysis Set

<< Programming note: Same shell as table 14.2-28.3 >>

Repeat for Immunophenotypically aberrant CD34 negative cells:

Table 14.2-31.1 Descriptive Statistics for Immunophenotypically aberrant CD34- cells: Percentage from total CD34+ cells – LSC sub-study Full Analysis Set

<< Programming note: Same shell as table 14.2-28.1 , exclude p-values >>

Table 14.2-31.2 Descriptive Statistics for number of events sorted in Immunophenotypically aberrant CD34-cells- LSC sub-study Full Analysis Set

<< Programming note: Same shell as table 14.2-28.1 , exclude p-values >>

Table 14.2-31.3 Ph+ by HIS status, in Immunophenotypically aberrant CD34- cells – LSC sub-study Full Analysis Set

<< Programming note: Same shell as table 14.2-28.3 >>

Table 14.2-31.4 Descriptive statistics of Ph+ in Immunophenotypically aberrant CD34- cells– LSC sub-study Full Analysis Set

<< Programming note: Same shell as table 14.2-28.1 , exclude p-values >>

Table 14.2-31.5 BCR-ABL by RT-PCR status, in Immunophenotypically aberrant CD34- cells – LSC sub-study Full Analysis Set

<< Programming note: Same shell as table 14.2-28.3 >>

#### By prior Imatinib treatment duration

## Table 14.2-32.1 Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase by duration of prior exposure to Imatinib - Full Analysis Set

Duration of prior exposure to Imatinib (years) < 2Duration of prior exposure to Imatinib (years) >= 2 to <5Duration of prior exposure to Imatinib (years) >= 5

| | Arm 1<br>N=xx | Arm 2<br>N=xx | Randomized<br>N=xx | Not Randomized N=xx | Total<br>N=xx |
|---|---|---|---|---|---|
| Molecular response 4.0 at baseline | | | | | |
| Number of responders | XX | XX | XX | XX | XX |
| Percentage (95% CI) | xx (xx.x,<br>xx.x) | xx (xx.x, xx.x) | xx (xx.x, xx.x) | xx (xx.x, xx.x) | xx (xx.x, xx.x) |
| Cumulative molecular response 4.0 up to 3 months (Day 91) Cumulative number of responders | xx | xx | xx | xx | xx |
| Cumulative percentage (95% CI) | xx (xx.x,<br>xx.x) | xx (xx.x, xx.x) | xx (xx.x, xx.x) | xx (xx.x, xx.x) | xx (xx.x, xx.x) |
| Cumulative molecular response 4.0 up to 6 months (Day 182) | | | | | |
| ••• | • • • | • • • | • • • | • • • | • • • |
| Repeat until 24 months | | | | | |
| Cumulative molecular response 4.0 up to 24 months (Day 730) | | | | | |
| Cumulative number of responders | XX | XX | XX | XX | XX |
| Cumulative percentage (95% CI) | xx (xx.x,<br>xx.x) | xx (xx.x, xx.x) | xx (xx.x, xx.x) | xx (xx.x, xx.x) | xx (xx.x, xx.x) |

<sup>-</sup> Percentage based on the number of patients included in the analysis population (N)

<sup>-</sup> Confidence Interval calculated as per Clopper-Pearson exact method.

### Table 14.2-32.1.1 Raw cumulative incidence of MMR during pre-randomization Induction/Consolidation phase by by prior Imatib treatment duration – LSC sub-study Full Analysis Set

<< Programming note: Same shell as table 14.2-32.1, for LSC sub-study FAS>>

## Table 14.2-32.2 Raw cumulative incidence of MMR during post-randomization consolidation phase (ARM 2) by prior Imatib treatment duration - Subset of Full Analysis Set, randomized to ARM 2

| Duration of prior exposure (years) < 2 Duration of prior exposure (years) >= 2 to <5 Duration of prior exposure (years) >= 5 | N=xx |
|---|---|
| Molecular response 4.0 at baseline | |
| Number of responders | XX |
| Percentage (95% CI) | xx (xx.x, xx.x) |
| Cumulative molecular response 4.0 up to 27 months (Day 822) Cumulative number of responders Cumulative percentage (95% CI) | xx<br>xx (xx.x, xx.x) |
| Cumulative molecular response 4.0 up to 30 months (Day 913) | |
| Depart while 26 months | • • • |
| Repeat until 36 months | |
| Cumulative molecular response 4.0 up to 36 months (Day 1096) | |
| Cumulative number of responders | XX |
| Cumulative percentage (95% CI) | xx (xx.x, xx.x) |

<sup>-</sup> Percentage based on the number of patients included in the analysis population (N)

<sup>-</sup> Confidence Interval calculated as per Clopper-Pearson exact method

# Table 14.2-32.2.1 Raw cumulative incidence of MMR during post-randomization consolidation phase (ARM 2) by prior lmatib treatment duration - Subset of LSC sub-study Full Analysis Set , randomized to ARM 2

<< Programming note: Same shell as table 14.2-32.2, for LSC sub-study FAS ARM 2>>

### Table 14.2-32.3 Raw cumulative incidence of MMR during re-treatment phase by prior lmatib treatment duration – Subset of Full Analysis Set entering the re-treatment phase

<< Programming note:

- Same shell as Table 14.2-32.1, but for re-treatment two arms >>

Add footnote: \*For month 27 onwards, only Arm1 patients considered for Total in percentages denominator." Programing note added."

Table 14.2-33.1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase by prior Imatib treatment duration - Full Analysis Set

<< Programming note: Same shell as table 14.2-32.1, for MR 4.0 >>

Table 14.2-33.1.1 Raw cumulative incidence of MR 4.0 during pre-randomization Induction/Consolidation phase by prior Imatib treatment duration – LSC sub-study Full Analysis Set

<< Programming note: Same shell as table 14.2-32.1.1, for MR 4.0 >>

Table 14.2-33.2 Raw cumulative incidence of MR 4.0 during post-randomization consolidation phase (ARM 2) by prior Imatib treatment duration - Subset of Full Analysis Set, randomized to ARM 2

<< Programming note: Same shell as table 14.2-32.2, for MR 4.0 >>

Table 14.2-33.2.1 Raw cumulative incidence of MR 4.0 during post-randomization consolidation phase (ARM 2) by prior lmatib treatment duration - Subset of LSC sub-study Full Analysis Set , randomized to ARM 2

<< Programming note: Same shell as table 14.2-32.2.1, for MR 4.0 >>

Table 14.2-33.3 Raw cumulative incidence of MR 4.0 during re-treatment phase by prior lmatib treatment duration – Subset of Full Analysis Set entering the re-treatment phase

<< Programming note: Same shell as table 14.2-32.3, for MR 4.0 >>
Add footnote: \*For month 27 onwards, only Arm1 patients considered for Total in percentages denominator." Programing note
added."

Table 14.2-34.1 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase by prior Imatib treatment duration - Full Analysis Set

<< Programming note: Same shell as table 14.2-32.1, for MR 4.5 >>

Table 14.2-34.1.1 Raw cumulative incidence of MR 4.5 during pre-randomization Induction/Consolidation phase by prior Imatib treatment duration – LSC sub-study Full Analysis Set

<< Programming note: Same shell as table 14.2-32.1.1, for MR 4.5 >>

Table 14.2-34.2 Raw cumulative incidence of MR 4.5 during post-randomization consolidation phase (ARM 2) by prior Imatib treatment duration - Subset of Full Analysis Set, randomized to ARM 2

<< Programming note: Same shell as table 14.2-32.2, for MR 4.5 >>

Table 14.2-34.2.1 Raw cumulative incidence of MR 4.5 during post-randomization consolidation phase (ARM 2) by prior lmatib treatment duration - Subset of LSC sub-study Full Analysis Set , randomized to ARM 2

<< Programming note: Same shell as table 14.2-32.2.1, for MR 4.5 >>

Table 14.2-34.3 Raw cumulative incidence of MR 4.5 during re-treatment phase by prior lmatib treatment duration – Subset of Full Analysis Set entering the re-treatment phase

<< Programming note: Same shell as table 14.2-32.3, for MR 4.5 >>
Add footnote: \*For month 27 onwards, only Arml patients considered for Total in percentages denominator." Programing note
added."

**Listings (Section 14.2)** 

### Section 14.3 - Safety data

### Figures (Section 14.3)

Not applicable.

### Tables (Section 14.3)

Table 14.3-1.1 Duration of exposure to study treatment during pre-randomization Induction/Consolidation—Safety Set

| | Arm 1 | Arm 2 | Randomized | Not Randomized | Total |
|---|---|---|---|---|---|
| | N=xx | N=xx | N=xx | N=xx | N=xx |
| Exposure (months) - n (%) | | | | | |
| < 6 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| >= 6 - < 12 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| >= 12 - < 18 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| >= 18 - < =24 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| > 24 | xx (xx.x) | | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Exposure (months) | | | | | |
| n | XX | Xx | Xx | Xx | XX |
| Mean | XX.X | xx.x | XX.X | XX.X | xx.x |
| SD | x.xx | X.XX | X.XX | X.XX | X.XX |
| 25th Percentile | XX.X | xx.x | XX.X | XX.X | xx.x |
| Median | XX.X | xx.x | XX.X | XX.X | xx.x |
| 75th Percentile | xx.x | XX.X | XX.X | XX.X | XX.X |
| Min-Max | xx.x- xx.x | xx.x- xx.x | xx.x- xx.x | xx.x- xx.x | xx.x- xx.x |

<sup>-</sup> Exposure (months) = (date of last administration - date of first administration in Induction/Consolidation phase + 1)/30.4375.

<sup>-</sup> Safety Set consists of all patients who received at least one dose of study drug, excluding patients with PD severity codes (0, 5, 8).

### Table 14.3-1.1.1 Duration of exposure to study treatment during pre-randomization Induction/Consolidation– LSC substudy Safety Set

<< Programming note: Same shell as table 14.3-1.1, for LSC sub-study SAF >>

## Table 14.3-1.2 Duration of exposure to study treatment during post-randomization Consolidation phase (ARM 2) - Subset of Safety Set randomized to Arm 2

<< Programming note: Same shell as table 14.3-1.1.1 with arm 2 only.
Use <6, >=6 to <=12 and >12 categories.
Footnote:
- Exposure (months) = (date of last administration - date of first administration in post-randomization consolidation phase +
1)/30.4375.
- Safety Set consists of all patients who received at least one dose of study drug, excluding patients with PD severity codes
(0, 5, 8).

## Table 14.3-1.2.1 Duration of exposure to study treatment during post-randomization Consolidation phase (ARM 2) - Subset of LSC sub-study Safety Set randomized to Arm 2

<< Programming note: Same shell as table 14.3-1.2, for LSC sub-study SAF >>

Table 14.3-1.1.3 Duration of exposure to study treatment during re-treatment phase – Subset of Safety Set entering the re-treatment phase

| J | Arm 1 | Arm 2 | Total |
|---------------------------|------------|------------|------------|
| | N=XX | N=xx | N=xx |
| Exposure (months) - n (%) | | | |
| < 6 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| >= 6 - < 12 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| >= 12 - < 18 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| >= 18 - < 24 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| >= 24 - < 30 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| >= 30 - < 36 | xx (xx.x) | | xx (xx.x) |
| >= 36 | xx (xx.x) | | xx (xx.x) |
| Exposure (months) | | | |
| n | XX | Xx | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | X.XX | X.XX | X.XX |
| 25th Percentile | XX.X | XX.X | XX.X |
| Median | XX.X | XX.X | XX.X |
| 75th Percentile | XX.X | XX.X | XX.X |
| Min-Max | xx.x- xx.x | xx.x- xx.x | xx.x- xx.x |

<sup>-</sup> Exposure (months) = (date of last administration - date of first administration in RT phase + 1)/30.4375.

Table 14.3-1.1.21 Duration of exposure to study treatment during pre-randomization Induction/Consolidation phase, by stable MR4.0 at 24 months and halving time - Safety Set

<sup>-</sup> Patients randomized to Arm 1 have 24 months of treatment and a maximum of 36 months of re-treatment.

<sup>-</sup> Patients randomized to Arm 2 have 36 months of treatment and a maximum of 24 months of re-treatment.

<sup>-</sup> Safety Set consists of all patients who received at least one dose of study drug, excluding patients with PD severity codes (0, 5, 8).

Halving time <= 3 months
Halving time > 3 months

| | Stable MR4.0 at Month 24 N=xx | | | Unstable MR4.0 at Month 24<br>N=xx | | Total<br>N=xx |
|---|---|---|---|---|---|---|
| | Randomized<br>N=xx | Not<br>Randomized<br>N=xx | Randomized<br>N=xx | Not<br>Randomized<br>N=xx | Randomized<br>N=xx | Not<br>Randomized<br>N=xx |
| Exposure (months) - n (%) | | | | | | |
| < 6 | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| >= 6 - < 12 | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| >= 12 - < 18 | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| >= 18 - <= 24 | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| > 24 | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Exposure (months) | | | | | | |
| n | xx | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | X.XX | X.XX | X.XX | x.xx | X.XX | X.XX |
| 25th Percentile | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| 75th Percentile | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min-Max | xx.x- xx.x | xx.x- xx.x | xx.x- xx.x | xx.x- xx.x | xx.x- xx.x | xx.x- xx.x |

<sup>-</sup> Exposure (months) = (date of last administration - date of first administration in Induction/Consolidation phase + 1)/30.4375.

<sup>-</sup> Safety Set consists of all patients who received at least one dose of study drug, excluding patients with PD severity codes (0, 5, 8).
### Table 14.3-1.1.22 Duration of exposure to study treatment during pre-randomization Induction/Consolidation phase, by stable MR4.0 by 24 months and halving time - Safety Set

Halving time <= 3 months
Halving time > 3 months

| , | | ) by Month 24<br>=xx | | 0 by Month 24<br>Exx | Total<br>N=xx | |
|---|---|---|---|---|---|---|
| | Randomized<br>N=xx | Not<br>Randomized<br>N=xx | Randomized<br>N=xx | Not<br>Randomized<br>N=xx | Randomized<br>N=xx | Not<br>Randomized<br>N=xx |
| Exposure (months) - n (%) | | | | | | |
| < 6 | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| >= 6 - < 12 | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| >= 12 - < 18 | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| >= 18 - <= 24 | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| > 24 | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Exposure (months) | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | xx.x | XX.X | XX.X |
| SD | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| 25th Percentile | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| 75th Percentile | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min-Max | xx.x- xx.x | xx.x- xx.x | xx.x- xx.x | xx.x- xx.x | xx.x- xx.x | xx.x- xx.x |

<sup>-</sup> Exposure (months) = (date of last administration - date of first administration in Induction/Consolidation phase + 1)/30.4375.

<sup>-</sup> Safety Set consists of all patients who received at least one dose of study drug, excluding patients with PD severity codes (0, 5, 8).

Table 14.3-2.1 Relative dose intensity and average daily dose during pre-randomization Induction/Consolidation phase – Safety Set

| | Arm 1 | Arm 2 | Randomized | Not Randomized | Total |
|---|---|---|---|---|---|
| | N=xx | N=xx | N=xx | N=xx | N=xx |
| Relative dose intensity | _ | | | | |
| n (%) | | | | | |
| < 70% | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| >=70 - <90% | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| >=90 - <100% | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| >=100% | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Relative dose intensity | | | | | |
| n | XX | XX | xx | XX | XX |
| Mean | xx.x | XX.X | xx.x | XX.X | XX.X |
| SD | x.xx | x.xx | x.xx | X.XX | X.XX |
| 25th Percentile | xx.x | XX.X | xx.x | XX.X | XX.X |
| Median | xx.x | XX.X | xx.x | XX.X | XX.X |
| 75th Percentile | xx.x | XX.X | xx.x | XX.X | XX.X |
| Min-Max | XX.X- XX.X | xx.x- xx.x | xx.x- xx.x | xx.x- xx.x | xx.x- xx.x |
| Average daily dose | | | | | |
| (mg/day) | | | | | |
| n | XX | XX | xx | XX | XX |
| Mean | xx.x | XX.X | xx.x | XX.X | XX.X |
| SD | x.xx | x.xx | x.xx | x.xx | X.XX |
| 25th Percentile | XX.X | XX.X | xx.x | XX.X | XX.X |
| Median | XX.X | xx.x | xx.x | XX.X | XX.X |
| 75th Percentile | XX.X | XX.X | xx.x | XX.X | XX.X |
| Min-Max | xx.x- xx.x | xx.x- xx.x | xx.x- xx.x | xx.x- xx.x | xx.x- xx.x |

<sup>-</sup> Actual dose intensity = Cumulative dose (mg) / Duration of exposure (day)

<sup>-</sup> Relative dose intensity = [Actual dose intensity /Planned dose intensity]\*100

<sup>-</sup> Average daily dose = Cumulative dose (mg) /  $(date\ of\ end\ of\ medication\ -\ date\ of\ start\ of\ medication\ +\ 1)$  (day) where number of drug free days are included in the denominator.

### Table 14.3-2.1.1 Relative dose intensity and average daily dose during pre-randomization Induction/Consolidation phase – LSC sub-study Safety Set

<< Programming note: Same shell as table 14.3-2.1, for LSC sub-study SAF >>

Table 14.3-2.2 Relative dose intensity and average daily dose during post-randomization consolidation phase (ARM 2) – Subset of Safety Set randomized to Arm 2

<< Programming note: Same shell as table 14.3-1.2.1 with arm 2 only.</pre>

Table 14.3-2.2.1 Relative dose intensity and average daily dose during post-randomization consolidation phase (ARM 2) – Subset of LSC sub-study Safety Set randomized to Arm 2

<< Programming note: Same shell as table 14.3-2.2, for LSC sub-study SAF ARM 2 only >>

Table 14.3-2.3 Relative dose intensity and average daily dose during re-treatment phase – Subset of Safety Set entering the re-treatment phase

| got onto mg mo | Arm 1 | Arm 2 | Total |
|-----------------------------|------------|------------|------------|
| | N=XX | N=XX | N=xx |
| Relative dose intensity - n | (%) | | |
| < 70% | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| >=70 - <90% | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| >=90 - <100% | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| >=100% | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Relative dose intensity | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | X.XX | X.XX | X.XX |
| 25th Percentile | XX.X | XX.X | XX.X |
| Median | XX.X | XX.X | XX.X |
| 75th Percentile | XX.X | XX.X | XX.X |
| Min-Max | xx.x- xx.x | xx.x- xx.x | xx.x- xx.x |
| Average daily dose (mg/day) | | | |
| n | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X |
| SD | X.XX | X.XX | X.XX |
| 25th Percentile | XX.X | XX.X | XX.X |
| Median | XX.X | XX.X | XX.X |
| 75th Percentile | XX.X | XX.X | XX.X |
| Min-Max | xx.x- xx.x | xx.x- xx.x | xx.x- xx.x |

<sup>-</sup> Actual dose intensity = Cumulative dose (mg) / Duration of exposure (day)

<sup>-</sup> Relative dose intensity = [Actual dose intensity /Planned dose intensity]\*100

<sup>-</sup> Average daily dose = Cumulative dose (mg) / (date of end of medication - date of start of medication + 1) (day) where number of drug free days are included in the denominator

Table 14.3-3.1 Dose reduction and interruption during pre-randomization Induction/Consolidation phase - Safety Set

| | Arm 1<br>N=xx | Arm 2<br>N=xx | Randomized<br>N=xx | Not Randomized<br>N=xx | Total<br>N=xx |
|---|---|---|---|---|---|
| Number of reductions / interruptions | | | | | |
| • | | | | | |
| 0 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2-3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| >=4 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of patients with at least one dose reduction/interruption by reason | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Adverse event | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Dosing error | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Lab test abnormality | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Scheduling conflict | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Missing | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

<sup>-</sup> A patient with multiple occurrences of a reason for dose reduction or interruption is only counted once in that category.

Table 14.3-3.1.1 Dose reduction and interruption during pre-randomization Induction/Consolidation phase – LSC sub-study Safety Set

<sup>-</sup> A patient with multiple reasons for dose reduction or interruption is only counted once in the total row.

<sup>-</sup> Percentage based on the number of patients included in the analysis population (N).

# Table 14.3-3.2 Dose reduction and interruption during post-randomization consolidation phase (ARM 2) – Subset of Safety Set randomized to Arm 2

<< Programming note: Same shell as table 14.3-1.3.1 with arm 2 only.</pre>

Add following footnote as first:

- All medication starting at or after first study treatment exposure and before-randomization are reported in this table during the post-randomization consolidation phase.

#### Add footnote:

- 15 patients from ARM 2 discontinued during post-Randomization Consolidation phase.

### Table 14.3-3.2.1 Dose reduction and interruption during post-randomization consolidation phase (ARM 2) – Subset of LSC sub-study Safety Set randomized to Arm 2

<< Programming note: Same shell as table 14.3-3.2, for LSC sub-study SAF >>

Table 14.3-3.3 Dose reduction and interruption during re-treatment phase – Subset of Safety Set entering the re-treatment phase

| | Arm 1<br>N=xx | Arm 2<br>N=xx | Total<br>N=xx |
|---|---|---|---|
| Number of reductions / interruptions | | | |
| 0<br>1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2-3 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| >=4 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of patients with at least one dose reduction/interruption by reason | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Adverse event | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Dosing error | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Lab test abnormality | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Scheduling conflict | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Missing | xx (xx.x) | xx (xx.x) | xx (xx.x) |

<sup>-</sup> A patient with multiple occurrences of a reason for dose reduction or interruption is only counted once in that category.

<sup>-</sup> A patient with multiple reasons for dose reduction or interruption is only counted once in the total row.

<sup>-</sup> Percentage based on the number of patients included in the analysis population (N).

Table 14.3-4.1 Concomitant medication by ATC class and preferred term during pre-randomization Induction/Consolidation phase Full Analysis Set

| | Arm 1<br>N=xx | Arm 2<br>N=xx | Randomized<br>N=xx | Not<br>randomized<br>N=xx | Total<br>N=xx |
|---|---|---|---|---|---|
| Any ATC class<br>-Total | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ATC class 1 | | | | | |
| -Total | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred term 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred term 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ATC class 2 | | | | | |
| -Total | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred term 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred term 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

<sup>-</sup> All medication starting at or after enrollment and before randomization or DBL date or study completion/discontinuation are reported in this table.

Table 14.3-4.1.1 Concomitant medication by ATC class and preferred term during pre-randomization Induction/Consolidation phase LSC sub-study Full Analysis Set

<sup>-</sup> ATC classes are presented alphabetically; preferred terms are sorted within ATC class by frequency.

<sup>-</sup> A medication can appear with more than one ATC class.

<sup>-</sup> A patient with multiple occurrences of a PT is counted only once in the PT class.

<sup>-</sup> A patient with multiple PT within an ATC class is counted only once in the row describing the ATC class.

<sup>-</sup> Percentage based on the number of patients included in the analysis population (N).

Table 14.3-4.2 Concomitant medication by ATC class and preferred term during post-randomization consolidation phase (ARM 2)— Subset of Full Analysis Set randomized to Arm 2

| | N=xx |
|---|---|
| Any ATC class -Total | xx (xx.x) |
| ATC class 1 -Total Preferred term 1 Preferred term 2 | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) |
| ATC class 2 -Total Preferred term 1 Preferred term 2 | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) |
| Etc. | |

<sup>-</sup> All medication starting during the post-randomization consolidation phase.

#### << Programming notes:

All data from CMD must be taken after checking the start date is not before date of Visit 1. Note that an edit check is performed by Data Management to check that the starting date is not before Date of visit 1.

Select DTAREP1C=1 (Is there any data to be reported? = yes) and CMDTYP1C=3 (Concomitant medication)

If ATC2 is missing and PT\_TXT is not missing, then set "NON DRUG, THERAPIES and PROCEDURES" to ATC class

>>

<sup>-</sup> ATC classes are presented alphabetically; preferred terms are sorted within ATC class by frequency.

<sup>-</sup> A medication can appear with more than one ATC class.

<sup>-</sup> A patient with multiple occurrences of a PT is counted only once in the PT class.

<sup>-</sup> A patient with multiple PT within an ATC class is counted only once in the row describing the ATC class.

<sup>-</sup> Percentage based on the number of patients included in the analysis population (N).

Table 14.3-4.2.1 Concomitant medication by ATC class and preferred term during post-randomization consolidation phase (ARM 2)— Subset of LSC sub-study Full Analysis Set randomized to Arm 2

<< Programming note: Same shell as table 14.3-2, for LSC sub-study FAS >>

Table 14.3-4.3 Concomitant medication by ATC class and preferred term during TFR phase – Subset of Full Analysis Set entering the TFR phase

| | Arm 1<br>N=xx | Arm 2<br>N=xx | Total<br>N=xx |
|-------------------------|---------------|---------------|---------------|
| Any ATC class<br>-Total | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ATC class 1 | | | |
| -Total | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred term 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred term 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ATC class 2 | | | |
| -Total | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred term 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred term 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |

<sup>-</sup> All medication starting at or after randomization and before the end of TFR phase or DBL date or study completion/discontinuation are reported in this table.

<sup>-</sup> ATC classes are presented alphabetically; preferred terms are sorted within ATC class by frequency.

<sup>-</sup> A medication can appear with more than one ATC class.

<sup>-</sup> A patient with multiple occurrences of a PT is counted only once in the PT class.

<sup>-</sup> A patient with multiple PT within an ATC class is counted only once in the row describing the ATC class.

<sup>-</sup> Patients randomized to Arm 1 have a maximum of 36 months of TFR phase; Patients randomized to Arm 2 have a maximum of 24 months of TFR phase.

<sup>-</sup> Percentage based on the number of patients included in the analysis population (N).

### Table 14.3-4.4 Concomitant medication by ATC class and preferred term during re-treatment phase – Subset of Full Analysis Set entering the re-treatment phase

<< Programming note: Same shell as table 14.3-4 .3 but on re-treatment phase. Display the first following footnote:

- All medication starting at or after start of re-treatment phase and before the DBL date or study completion/discontinuation are reported in this table.
- ATC classes are presented alphabetically; preferred terms are sorted within ATC class alphabetically.
- A medication can appear with more than one ATC class.

>>

- A patient with multiple occurrences of a PT is counted only once in the PT class.
- A patient with multiple PT within an ATC class is counted only once in the row describing the ATC class.
- Patients randomized to Arm 1 have 24 months of treatment and a maximum of 36 months of re-treatment.
  - Patients randomized to Arm 2 have 36 months of treatment and a maximum of 24 months of re-treatment.
- Percentage based on the number of patients included in the analysis population (N).

Table 14.3-5.1.1 Hematology shift table based on CTCAE grade during Pre-Randomization pre-randomization Induction/Consolidation –Full Analysis Set

| | | _Baseline | Ind/Cons_ | | Wo | rst v | alue du | | | domiz | ation I | nd/Co | ons treat | tment |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | Gr | rade 0 | Gr | rade 1 | Gı | rade 2 | Gr | ade 3 | G | rade 4 | Missing |
| Treatment | | | n | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n |
| | | Grade 0 | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| Arm 1 | | Grade 1 | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| (N=xxx) | | Grade 2 | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| | etc. | • | | | | | | | | | | | | |
| | | Missing | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| | | Total | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| | | Grade 0 | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | xx |
| Arm 2 | | Grade 1 | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| (N=xxx) | | Grade 2 | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| | etc. | | | | | | | | | | | | | |
| | | Missing | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| | | Total | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| | | Grade 0 | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | xx |
| Randomized | | Grade 1 | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| (N=xxx) | | • • • | • • | | | | | • • • | | | | • | • • | • • |
| | | Grade 0 | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | xx |
| Not Randomized | | Grade 1 | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| (N=xxx) | | • • • | • • | | | | | • • • | | | | • | • • | • • |
| | | Grade 0 | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | xx |
| Total | | Grade 1 | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| (N=xxx) | | Grade 2 | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| | etc. | • | | | | | | | | | | | | |
| | | Missing | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| | | Total | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |

<sup>-</sup> Baseline Ind/Cons corresponds to the last assessment before or on the first day of nilotinib intake during induction/consolidation phase.

#### NovartisConfidentialPage 288RAP Module 7.16-May-2021 (14:35)Protocol No CAMN107AIC0

- Percentage calculated by row, based on number of available patients at Baseline Ind/Cons with corresponding grade and at least one non-missing post baseline value.
- Grades as per CTCAE v 4.03.
- Grade 0 = Non-missing value below Grade 1.
- Laboratory assessments performed outside of re-treatment phase are not described.
- Patients randomized to Arm 1 have 24 months of treatment and a maximum of 36 months of re-treatment.
  - Patients randomized to Arm 2 have 36 months of treatment and a maximum of 24 months of re-treatment.

#### << Programming note:

- List of hematology parameters which have CTCAE grade in version 4.03 and have to be displayed: WBCs, absolute lymphocytes, absolute neutrophils, hemoglobin and platelets.
- Note that the scheduled and unscheduled records are considered in this summary.
- Do not display a line if all the records are 0 e.g. if there are no grade 4 at baseline the grade 4 line should not appear in the table.
- % calculated by row excluding the patients with missing post baseline.
- Note that a patient with Baseline only would be counted in the baseline count but would appear post baseline as missing and therefore would not be included in the denominator for the % calculation. >>

### Table 14.3-5.1.2 Hematology shift table based on CTCAE grade during post-randomization consolidation phase (ARM 2)– Subset of Full Analysis Set randomized to Arm 2

Parameter: xxxxx

| | | Base | line | | Worst on-treatment value | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | <del></del> | | | | Gr | rade 1 | Grade 2 | | Grade 3 | | Grade 4 | | Missing |
| | | | n | n | (%) | n | (응) | n | (%) | n | (응) | n | (%) | n |
| | | Grade 0 | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| | Grade | 1 xx | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | ζ |
| (N=xxx) | | Grade 2 | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| | etc. | | | | | | | | | | | | | |
| | | Missing | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| | | Total | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |

- Baseline is defined as the last assessment before or at the date the patient Randomized.
- Percentage calculated by row, based on number of available patients at Baseline with corresponding grade and at least one non-missing post baseline value.
- Grades as per CTCAE v 4.03.
- Grade 0 = Non-missing value below Grade 1.
- Laboratory assessments performed outside of post-randomization consolidation phase are not described.
- Patients randomized to Arm 2 have 12 months of treatment post-randomization and a maximum of 24 months of re-treatment.

#### << Programming note:

- List of hematology parameters which have CTCAE grade in version 4.03 and have to be displayed: WBCs, absolute lymphocytes, absolute neutrophils, hemoglobin and platelets.
- Note that the scheduled and unscheduled records are considered in this summary.
- Do not display a line if all the records are 0 e.g. if there are no grade 4 at baseline the grade 4 line should not appear in the table.
- % calculated by row excluding the patients with missing post baseline.
- Note that a patient with Baseline only would be counted in the baseline count but would appear post baseline as missing and therefore would not be included in the denominator for the % calculation. >>

Table 14.3-5.1.3 Hematology shift table based on CTCAE grade during re-treatment phase – Subset of Full Analysis Set entering the re-treatment phase

| | | Baseline | | Worst value during re-treatment | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | _ | | | Gr | ade 0 | Gı | ade 1 | Gr | cade 2 | Gr | cade 3 | Gı | cade 4 | Missing |
| Treatment | | | n | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n |
| | | Grade 0 | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| Arm 1 | | Grade 1 | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| (N=xxx) | | Grade 2 | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| | etc. | | | | | | | | | | | | | |
| | | Missing | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| | | Total | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| | | Grade 0 | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| Arm 2 | | Grade 1 | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| (N=xxx) | | Grade 2 | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| | etc. | | | | | | | | | | | | | |
| | | Missing | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| | | Total | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| | | Grade 0 | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| Total | | Grade 1 | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| (N=xxx) | | Grade 2 | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| | etc. | | | | | | | | | | | | | |
| | | Missing | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| | | Total | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |

<sup>-</sup> Baseline RT corresponds to the last assessment before or at the date the patient entered re-treatment phase.

Patients randomized to Arm 2 have 36 months of treatment and a maximum of 24 months of re-treatment.

<sup>-</sup> Percentage calculated by row, based on number of available patients at Baseline RT with corresponding grade and at least one non-missing post baseline value.

<sup>-</sup> Grades as per CTCAE v 4.03.

<sup>-</sup> Grade 0 = Non-missing value below Grade 1.

<sup>-</sup> Laboratory assessments performed outside of re-treatment phase are not described.- Patients randomized to Arm 1 have 24 months of treatment and a maximum of 36 months of re-treatment.

#### << Programming note:

- List of hematology parameters which have CTCAE grade in version 4.03 and have to be displayed: WBCs, absolute lymphocytes, absolute neutrophils, hemoglobin and platelets.
- Note that the scheduled and unscheduled records are considered in this summary.
- Do not display a line if all the records are 0 e.g. if there are no grade 4 at baseline the grade 4 line should not appear in the table.
- % calculated by row excluding the patients with missing post baseline.
- Note that a patient with Baseline only would be counted in the baseline count but would appear post baseline as missing and therefore would not be included in the denominator for the % calculation. >>

Table 14.3-5.1.4 Hematology shift table based on CTCAE grade during whole study period – Full Analysis Set

| | | Baseline | | | Worst value during whole study period | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | _ | | | Gı | Grade 0 | | ade 1 | Gi | rade 2 | Gı | rade 3 | Grade 4 | | Missing |
| Treatment | | | n | n | (응) | n | (%) | n | (%) | n | (응) | n | (%) | n |
| | | Grade 0 | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| Arm 1 | | Grade 1 | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| (N=xxx) | | Grade 2 | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| | etc. | | | | | | | | | | | | | |
| | | Missing | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| | | Total | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| | | Grade 0 | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| Arm 2 | | Grade 1 | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| (N=xxx) | | Grade 2 | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| | etc. | | | | | | | | | | | | | |
| | | Missing | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| | | Total | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| | | Grade 0 | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| Randomized | | Grade 1 | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| (N=xxx) | | • • • | • • | • • | | | | • • | • | • • | | | | • • |
| | | Grade 0 | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| Not Randomized | | Grade 1 | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| (N=xxx) | | • • • | • • | • • | | | | • • | • | • • | | • • | | • • |
| | | Grade 0 | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| Total | | Grade 1 | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| (N=xxx) | | Grade 2 | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| • | etc. | | | | • | | • | | , | | , | | - | |
| | | Missing | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| | | Total | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |

<sup>-</sup> Baseline is defined as the last available assessment before or at date of start of study treatment.

<sup>-</sup> Percentage calculated by row, based on number of available patients at Baseline with corresponding grade and at least one non-missing post baseline value.

- Grades as per CTCAE v 4.03.
- Grade 0 = Non-missing value below Grade 1.
- Laboratory assessments performed outside of study period are not described.
- Patients randomized to Arm 1 have 24 months of treatment and a maximum of 36 months of re-treatment.
  - Patients randomized to Arm 2 have 36 months of treatment and a maximum of 24 months of re-treatment.

#### << Programming note:

- List of hematology parameters which have CTCAE grade in version 4.03 and have to be displayed: WBCs, absolute lymphocytes, absolute neutrophils, hemoglobin and platelets.
- Note that the scheduled and unscheduled records are considered in this summary.
- Do not display a line if all the records are 0 e.g. if there are no grade 4 at baseline the grade 4 line should not appear in the table.
- % calculated by row excluding the patients with missing post baseline.
- Note that a patient with Baseline only would be counted in the baseline count but would appear post baseline as missing and therefore would not be included in the denominator for the % calculation. >>

### Table 14.3-5.1.5 Hematology shift table based on CTCAE grade during re-treatment phase, SDV sensitivity – Subset of Full Analysis Set entering the re-treatment phase

<< Programming note: Same shell as Table 14.3-5.1.3, for SDV sensitivity analysis>>
Add footnote:

- SDV sensitivity: Excluding patient visits involved in SDV issues during final data review due to COVID-19.

#### Table 14.3-5.1.6 Hematology shift table based on CTCAE grade during whole study period , SDV sensitivity– Full Analysis Set

<< Programming note: Same shell as Table 14.3-5.1.4, for SDV sensitivity analysis>> Add footnote:

- SDV sensitivity: Excluding patient visits involved in SDV issues during final data review due to COVID-19.

### Table 14.3-5.2.1 Biochemistry shift table based on CTCAE grade during post-randomization consolidation phase (ARM 2)— Subset of Full Analysis Set randomized to Arm 2

<< Programming note: Same shell as table 14.3-5.1.2 >>

- List of biochemistry parameters which have CTCAE grade in version 4.03 and have to be displayed: bilirubin (total, indirect and direct), aspartate aminotransferase (AST), alanine aminotransferase (ALT), sodium (hyper & hypo), potassium (hyper & hypo), calcium (hyper & hypo), magnesium (hyper & hypo), glucose (hyper & hypo), creatinine, phosphate (or serum phosphorus), lipase, amylase, total cholesterol and triglycerides.
- Note that for bi-directional parameters (where hyper and hypo abnormalities are defined), the value graded in the other direction (hyper if the parameter of interest is hypo) is counted as a grade 0. Note that the scheduled and unscheduled records are considered in this summary. Make sure the parameters to display can be changed, added and removed easily. >>

#### Table 14.3-5.2.2 Biochemistry shift table based on CTCAE grade during re-treatment phase— Subset of Full Analysis Set entering the re-treatment phase

<< Programming note: Same shell as table 14.3-5.1.3 >>

Table 14.3-5.2.3 Biochemistry shift table based on CTCAE grade during whole study period – Full Analysis Set << Programming note: Same shell as table 14.3-5.1.4 >>

#### Table 14.3-5.2.4 Biochemistry shift table based on CTCAE grade during re-treatment phase, SDV sensitivity—Subset of Full Analysis Set entering the re-treatment phase

<< Programming note: Same shell as Table 14.3-5.2.2, for SDV sensitivity analysis>> Add footnote:

- SDV sensitivity: Excluding patient visits involved in SDV issues during final data review due to COVID-19.

#### Table 14.3-5.2.5 Biochemistry shift table based on CTCAE grade during whole study period, SDV sensitivity – Full Analysis Set

<< Programming note: Same shell as Table 14.3-5.2.3, for SDV sensitivity analysis>>
Add footnote:

- SDV sensitivity: Excluding patient visits involved in SDV issues during final data review due to COVID-19.

Table 14.3-6.1.1 Hematology shift table based on normal range for parameters with no defined CTCAE grades during post-randomization consolidation phase (ARM 2)– Subset of Full Analysis Set randomized to Arm 2

| | | | | _ Wc | rst va | lue d | luring p | post- | random | izati | on cons | olidation |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Basel: | ine | I | WOL | No | rmal | F | Iigh | Higl | n & Low | Missing |
| Treatment | | | n | n | (%) | n | (%) | n | (%) | n | (%) | n |
| (N=xxx) | Low | xx<br>Normal<br>High<br>Missing | XX<br>XX<br>XX | XX | xx (:<br>(xx.x)<br>(xx.x)<br>(xx.x) | XX | xx (:<br>(xx.x)<br>(xx.x)<br>(xx.x) | XX | (xx.x) | XX | xx<br>(xx.x)<br>(xx.x)<br>(xx.x) | xx<br>xx<br>xx |
| | | Total | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |

<sup>-</sup>Baseline is defined as the last assessment before or at the date the patient Randomized.

<<pre><<Pre>rogramming note: List of Hematology parameters which do not have CTCAE grade in version 4.03 and have to be displayed:
eosinophils, basophils, monocytes, promyelocytes, myelocytes, metamyelocytes and blast.

Do not display a line if all the records are 0.

>>

Note that a patient with Baseline only would be counted in the baseline count but would appear post baseline as missing and therefore would not be included in the denominator for the % calculation.

<sup>-</sup> Percentage calculated by row, based on number of available patients at Baseline with corresponding level and at least one non-missing post baseline value. Low/High categories defined by normal ranges.

<sup>-</sup> High & Low category defined when patients experienced low and high values (they are not count in Low category or High category). Only parameters without CTCAE grades are included.

<sup>-</sup> Laboratory assessments performed outside of the post-randomization consolidation phase are not described.

<sup>-</sup> Patients randomized to Arm 2 have 12 months of treatment post-randomization and a maximum of 24 months of re-treatment.

<sup>%</sup> calculated by row excluding the patients with missing post baseline.

Table 14.3-6.1.2 Hematology shift table based on normal range for parameters with no defined CTCAE grades during re-treatment phase – Subset of Full Analysis Set entering the re-treatment phase

| | | | | V | Vorst | value | duri | .ng re-t | treat | tment | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Baseline | RT | _ I | WO | No | ormal | F | Iigh | Hig | gh & Low | Missing |
| Treatment | | n | n | (%) | n | (용) | n | (%) | n | (%) | n |
| Arm 1 | Low | XX | XX | (xx.x) | xx | (xx.x) | XX | (xx.x) | xx | (xx.x) | XX |
| (N=xxx) | Normal | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| | High | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| | Missing | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| | Total | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| Arm 2 | Low | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| (N=xxx) | Normal | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| | High | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| | Missing | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| | Total | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| Total | Low | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| (N=xxx) | Normal | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| | High | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| | Missing | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| | Total | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |

<sup>-</sup> Baseline RT corresponds to the last assessment before or at the date the patient entered re-treatment phase.

<sup>-</sup> Percentage calculated by row, based on number of available patients at Baseline RT with corresponding level and at least one non-missing post baseline value. Low/High categories defined by normal ranges.

<sup>-</sup> High & Low category defined when patients experienced low and high values (they are not count in Low category or High category). Only parameters without CTCAE grades are included.

<sup>-</sup> Laboratory assessments performed outside of re-treatment phase are not described.

<sup>-</sup> Patients randomized to Arm 1 have 24 months of treatment and a maximum of 36 months of re-treatment.

<sup>-</sup> Patients randomized to Arm 2 have 36 months of treatment and a maximum of 24 months of re-treatment.

Table 14.3-6.1.3 Hematology shift table based on normal range for parameters with no defined CTCAE grades during whole study period –Full Analysis Set

| | | | | | | | - | whole | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Baseline_ | | Low | | Norma | | High | | igh 8 | | Missing |
| Treatment | | n | n | (%) | n | (%) | n | (%) | n | (%) | n |
| Arm 1 | Low | xx | ×× | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| (N=xxx) | Normal | XX | XX | (xx.x) | XX | (xx.x) | xx | (xx.x) | | (xx.x) | |
| , | High | XX | XX | (xx.x) | | (xx.x) | | (xx.x) | | (xx.x) | |
| | Missing | XX | XX | (xx.x) | | (xx.x) | | (xx.x) | | (xx.x) | |
| | Total | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| Arm 2 | Low | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | xx |
| (N=xxx) | Normal | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| | High | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| | Missing | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| | Total | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| Randomized | Low | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| (N=xxx) | Normal | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| | High | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| | Missing | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| | Total | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| Not Randomized | Low | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| (N=xxx) | Normal | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| | High | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| | Missing | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| | Total | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| Total | Low | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | xx | (xx.x) | XX |
| (N=xxx) | Normal | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| | High | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| | Missing | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| | Total | XX | XX | (xx.x) | XX | (xx.x) | xx | (xx.x) | XX | (xx.x) | xx |

- Baseline is defined as the last available assessment before or at date of start of study treatment.
- Percentage calculated by row, based on number of available patients at Baseline with corresponding level and at least one non-missing post baseline value. Low/High categories defined by normal ranges.
- High & Low category defined when patients experienced low and high values (they are not count in Low category or High category). Only parameters without CTCAE grades are included.
- Laboratory assessments performed outside of study period are not described.
- Patients randomized to Arm 1 have 24 months of treatment and a maximum of 36 months of re-treatment.
  - Patients randomized to Arm 2 have 36 months of treatment and a maximum of 24 months of re-treatment.

# Table 14.3-6.1.4 Hematology shift table based on normal range for parameters with no defined CTCAE grades during re-treatment phase, SDV sensitivity – Subset of Full Analysis Set entering the re-treatment phase

<< Programming note: Same shell as Table 14.3-6.1.2, for SDV sensitivity analysis>> Add footnote:

- SDV sensitivity: Excluding patient visits involved in SDV issues during final data review due to COVID-19.

# Table 14.3-6.1.5 Hematology shift table based on normal range for parameters with no defined CTCAE grades during whole study period, SDV sensitivity –Full Analysis Set

<< Programming note: Same shell as Table 14.3-6.1.3, for SDV sensitivity analysis>> Add footnote:

- SDV sensitivity: Excluding patient visits involved in SDV issues during final data review due to COVID-19.

Table 14.3-6.2.1 Biochemistry shift table based on normal range for parameters with no defined CTCAE grades during post-randomization consolidation phase (ARM 2) – Subset of Full Analysis Set randomized to Arm 2

<< Programming note: Same shell as table 14.3-6.1.1 >>

Table 14.3-6.2.2 Biochemistry shift table based on normal range for parameters with no defined CTCAE grades during re-treatment phase – Subset of Full Analysis Set entering the re-treatment phase <</pre>
<< Programming note: Same shell as table 14.3-6.1.2 >>

<< Programming note: Same shell as table 14.3-6.1.2 >>

Table 14.3-6.2.3 Biochemistry shift table based on normal range for parameters with no defined CTCAE grades during whole study period –Full Analysis Set

<< Same shell as table 14.3-6.1.3 >>

Table 14.3-6.2.4 Biochemistry shift table based on normal range for parameters with no defined CTCAE grades during re-treatment phase, SDV sensitivity – Subset of Full Analysis Set entering the re-treatment phase

<< Programming note: Same shell as Table 14.3-6.2.2, for SDV sensitivity analysis>> Add footnote:

- SDV sensitivity: Excluding patient visits involved in SDV issues during final data review due to COVID-19.

Table 14.3-6.2.5 Biochemistry shift table based on normal range for parameters with no defined CTCAE grades during whole study period, SDV sensitivity –Full Analysis Set

<< Programming note: Same shell as Table 14.3-6.2.3, for SDV sensitivity analysis>> Add footnote:

- SDV sensitivity: Excluding patient visits involved in SDV issues during final data review due to COVID-19.

Table 14.3-7.1 ECG shift table based on notable values during Pre-randomization Induction Consolidation–Full Analysis Set

| | Parameter: QTcF (msec) | | | | | |
|---|---|---|---|---|---|---|
| | Baseline Ind/Cons | | Worst | on-treatment | value | |
| | | <=450 | >450 -480 | >480 - 500 | >500 | Missing |
| Treatment | n | n (%) | n (%) | n (%) | n (%) | n |
| | . 450 | , | , | , | , | |
| Arm 1 | <=450 xx | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX |
| (N=xxx) | >450 - 480 xx | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX |
| | >480 - 500 xx | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX |
| | >500 xx | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX |
| | Missing xx | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX |
| | Total xx | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX |
| Arm 2 | <=450 xx | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX |
| (N=xxx) | >450 - 480 xx | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX |
| , | >480 - 500 xx | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX |
| | >500 xx | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX |
| | Missing xx | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX |
| | Total xx | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX |
| | 4.50 | , | , | , | , | |
| Randomized | <=450 xx | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX |
| (N=xxx) | >450 - 480 xx | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX |
| | • | • • • | • • • | • • • | • • • | • • |
| Not Randomized | <=450 xx | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX |
| (N=xxx) | >450 - 480 xx | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX |
| | ••• | | | | | |
| Total | <=450 xx | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX |
| (N=xxx) | >450 - 480 xx | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX |
| (11-222) | | , , | , , | | , | |
| | <br>Total vv | ••• | ••• | ••• | ••• | • • |
| | Total xx | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX |

<sup>-</sup> Baseline Ind/Cons corresponds to the last assessment before or on the first day of nilotinib intake during induction/consolidation phase.

<sup>-</sup> Percentage for worst value is calculated by row, based on number of available patients at Baseline with corresponding category and at least one non-missing post baseline value.

<sup>-</sup> Unscheduled visits are included.

<sup>-</sup> Patients randomized to Arm 1 have 24 months of treatment and a maximum of 36 months of re-treatment.

<sup>-</sup> Patients randomized to Arm 2 have 36 months of treatment and a maximum of 24 months of re-treatment.

# Table 14.3-7.2 ECG shift table based on notable values during post-randomization consolidation phase (ARM 2) – Subset of Full Analysis Set randomized to Arm 2

| | | Par | ameter: QTcF (msec) | | |
|---|---|---|---|---|---|
| | Baseline | | Worst on-treatment v | <i>r</i> alue | |
| | <del></del> | <=450 | >450 -480 >480 - 500 | >500 | Missing |
| | n | n (%) | n (%) n (%) | n (%) | n |
| <=450 | xx xx (xx.x) | ( v.) | vv (vv v) vv (vv v) | 3737 | |
| | , , | xx (xx.x) | xx (xx.x) xx (xx.x) | XX | |
| (N=xxx) | >450 - 480 xx | xx (xx.x) | xx (xx.x) xx (xx.x) | xx (xx.x) | XX |
| | >480 - 500 xx | xx (xx.x) | xx (xx.x) xx (xx.x) | xx (xx.x) | XX |
| | >500 xx | xx (xx.x) | xx (xx.x) xx (xx.x) | xx (xx.x) | XX |
| | Missing xx | xx (xx.x) | xx (xx.x) xx (xx.x) | xx (xx.x) | XX |
| | Total xx | xx (xx.x) | xx (xx.x) xx (xx.x) | xx (xx.x) | XX |

- Baseline is defined as the last assessment before or at the date the patient Randomized.
- Percentage for worst value is calculated by row, based on number of available patients at Baseline with corresponding category and at least one non-missing post baseline value.
- Unscheduled visits are included.
- Patients randomized to Arm 2 have 12 months of treatment post-randomization and a maximum of 24 months of re-treatment.

<< Programming note: Only patients with all missing values post-baseline will be counted in the 'Missing' column.>>

Table 14.3-7.3 ECG shift table based on notable values during re-treatment phase – Subset of Full Analysis Set entering the re-treatment phase

| - | - | | | Par | ramet | er: QT | cF (m | sec) | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Baseline | RT | | | | Worst o | n-tre | atment v | value | | |
| | | | _< | =450 | >45 | 0 -480 | >480 | - 500 | > | 500 | Missing |
| Treatment | | n | n | (응) | n | (%) | n | (용) | n | (응) | n |
| Arm 1 | <=450 | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| (N=xxx) | >450 - 480 | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| | >480 - 500 | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| | >500 | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| | Missing | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| | Total | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| Arm 2 | <=450 | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| (N=xxx) | >450 - 480 | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| | >480 - 500 | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| | >500 | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| | Missing | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| | Total | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| Total | <=450 | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| (N=xxx) | >450 - 480 | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| | >480 - 500 | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| | >500 | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| | Missing | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |
| | Total | XX | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) | XX |

<sup>-</sup> Baseline RT corresponds to the last assessment before or at the date the patient entered re-treatment phase.

<<Pre><<Pre>rogramming note: Only patients with all missing values post-baseline will be counted in the 'Missing' column.>>

<sup>-</sup> Percentage for worst value is calculated by row, based on number of available patients at Baseline with corresponding category and at least one non-missing post baseline value.

<sup>-</sup> Unscheduled visits are included.

<sup>-</sup> Patients randomized to Arm 1 have 24 months of treatment and a maximum of 36 months of re-treatment.

<sup>-</sup> Patients randomized to Arm 2 have 36 months of treatment and a maximum of 24 months of re-treatment.

#### Table 14.3-7.4 Notable ECG values during pre-randomization Ind/Cons –Full Analysis Set

| | Arm 1 | Arm 2 | Randomized | Not Randomized | Total |
|---|---|---|---|---|---|
| | N=xx | N=xx | N=xx | N=xx | N=xx |
| | n (%) | n (%) | n (%) | n (%) | n (%) |
| QTcF (msec) | n=xx | n=xx | n=xx | n=xx | n=xx |
| <pre>Increase from baseline Ind/Cons &gt; 30 Increase from baseline Ind/Cons &gt; 60</pre> | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

<sup>-</sup> n is the number of patients meeting the criteria at least once.

<< Programming note: Patients can be included in multiple rows.>>

<sup>-</sup> Baseline Ind/Cons corresponds to the last assessment before or on the first day of nilotinib intake during induction/consolidation phase.

<sup>-</sup> Change from baseline: post baseline - baseline.

<sup>-</sup> Unscheduled visits are included.

<sup>-</sup> Percentage based on the number of patients with available data (n).

<sup>-</sup> Patients randomized to Arm 1 have 24 months of treatment and a maximum of 36 months of re-treatment.

<sup>-</sup> Patients randomized to Arm 2 have 36 months of treatment and a maximum of 24 months of re-treatment.

# Table 14.3-7.5 Notable ECG values during post-randomization consolidation phase (ARM 2)– Subset of Full Analysis Set randomized to Arm 2

| | N=xx |
|-----------------------------|-----------|
| | n (%) |
| QTcF (msec) | U=XX |
| Increase from baseline > 30 | xx (xx.x) |
| Increase from baseline > 60 | xx (xx.x) |

- n is the number of patients meeting the criteria at least once.
- Baseline is defined as the last assessment before or at the date the patient Randomized.
- Change from baseline: post baseline baseline.
- Unscheduled visits are included.
- Percentage based on the number of patients with available data (n).
- Patients randomized to Arm 2 have 12 months of treatment post-randomization and a maximum of 24 months of re-treatment.

<<pre><<Programming note: Patients can be included in multiple rows.>>

#### Table 14.3-7.6 Notable ECG values during re-treatment phase – Subset of Full Analysis Set entering the retreatment phase

| | Arm 1 | Arm 2 | Total |
|---|---|---|---|
| | N=xx | N=xx | N=xx |
| | n (%) | n (%) | n (%) |
| QTcF (msec) | n=xx | n=xx | n=xx |
| <pre>Increase from baseline RT &gt; 30 Increase from baseline RT &gt; 60</pre> | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | xx (xx.x) | xx (xx.x) | xx (xx.x) |

<sup>-</sup> n is the number of patients meeting the criteria at least once.

<< Programming note: Patients can be included in multiple rows.>>

#### Table 14.3-7.7 ECG shift table based on notable values during re-treatment phase, SDV sensitivity – Subset of Full Analysis Set entering the re-treatment phase

<< Programming note: Same shell as Table 14.3-7.3, for SDV sensitivity analysis>>
Add footnote:

- SDV sensitivity: Excluding patient visits involved in SDV issues during final data review due to COVID-19.

# Table 14.3-7.8 Notable ECG values during re-treatment phase, SDV sensitivity – Subset of Full Analysis Set entering the re-treatment phase

<< Programming note: Same shell as Table 14.3-7.6, for SDV sensitivity analysis>> Add footnote:

<sup>-</sup> Baseline RT is defined as the last available assessment before or at date of re-start of study treatment.

<sup>-</sup> Change from baseline: post baseline - baseline.

<sup>-</sup> Unscheduled visits are included.

<sup>-</sup> Percentage based on the number of patients with available data (n).

<sup>-</sup> Patients randomized to Arm 1 have 24 months of treatment and a maximum of 36 months of re-treatment.

<sup>-</sup> Patients randomized to Arm 2 have 36 months of treatment and a maximum of 24 months of re-treatment.

<sup>-</sup> SDV sensitivity: Excluding patient visits involved in SDV issues during final data review due to COVID-19

Table 14.3-8.1 Echocardiography assessment at baseline – Full Analysis Set

| | Arm 1<br>N=xxx<br>n (%) | Arm 2<br>N=xxx<br>n (%) | Randomized<br>N=xxx<br>n (%) | Not Randomized N=xxx n (%) | Total<br>N=xxx<br>n (%) |
|---|---|---|---|---|---|
| LVEF (%) | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | X.XX | X.XX | X.XX | X.XX | X.XX |
| 25th Percentile | XX.X | XX.X | XX.X | XX.X | XX.X |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| 75th Percentile | XX.X | XX.X | XX.X | xx.x | XX.X |
| Min-Max | xx.x - xx.x | xx.x - xx.x | xx.x - xx.x | xx.x - xx.x | xx.x - xx.x |
| Overall interpretation | n=xx | n=xx | n=xx | n=xx | n=xx |
| Normal | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Clinically insignificant abnormality | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Clinically significant abnormality | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

<sup>-</sup> Percentage based on the number of patients with available data (n)

Table 14.3-8.2 Echocardiography shift table based on overall interpretation - Full Analysis Set

| | Baseline | Worst post-baseline value | | | | |
|---|---|---|---|---|---|---|
| | | | | Clinic insign. | Clinic. sign. | |
| | | | Normal | abn. | abn. | Missing |
| Treatment | | n | n (%) | n (%) | n (%) | n |
| Arm 1 | Normal | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX |
| (N=xxx) | Clinic. insign. abn. | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX |
| | Clinic. sign. abn. | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX |
| | Missing | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX |
| | Total | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX |
| Arm 2 | Normal | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX |
| (N=xxx) | Clinic. insign. abn. | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX |
| | Clinic. sign. abn. | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX |
| | Missing | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX |
| | Total | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX |
| Randomized | Normal | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX |
| (N=xxx) | Clinic. insign. abn. | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX |
| | ••• | • • • | • • • | • • • | • • • | • • • |
| Not Randomized | Normal | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX |
| (N=xxx) | Clinic. insign. abn. | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX |
| | • • • | • • • | ••• | • • • | • • • | ••• |
| Total | Normal | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX |
| (N=xxx) | Clinic. insign. abn. | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX |
| | | | | | • • • | |

<sup>-</sup> Baseline is defined as the last available assessment before or at date of start of study treatment

Investigator's discretion if there are signs or symptoms of cardiotoxicity

<sup>-</sup> Percentage for worst value is calculated by row, based on number of available patients at Baseline with corresponding category and at least one non-missing post baseline value (1-24 months for Arm 1, Not Randomized and Total, 1-36 months for Arm 2).

<sup>-</sup> Unscheduled visits are included

<sup>-</sup> Clinic. insign abn. = Clinically insignificant abnormality, Clinic. sign. abn. = Clinically significant abnormality

<sup>-</sup> According to the protocol the Echocardiography is performed at screening and may be repeated at the

#### Table 14.3-8.3 Echocardiography shift table based on overall interpretation, SDV sensitivity - Full Analysis Set

<< Programming note: Same shell as Table 14.3-8.2, for SDV sensitivity analysis>> Add footnote:

- SDV sensitivity: Excluding patient visits involved in SDV issues during final data review due to COVID-19.

### Table 14.3-9.1 Summary statistics of total cholesterol, HDL, LDL, glucose, microalbumin and HbA1c over Induction/Consolidation phase – Full Analysis Set

All patients /Arm 1/ Arm 2/ /Randomized/ Not Randomized  $N{=}xx$ 

| Test (unit) | Visit | n | Mean | SD | 25 <sup>th</sup> Perc. | Median | 75 <sup>th</sup> Perc. | Missin |
|---|---|---|---|---|---|---|---|---|
| Total chole | sterol (mmol/L) | | | | | | | |
| | Screening | XX | X.XX | X.XX | X.XX | X.XX | X.XX | XX |
| | Baseline visit | XX | X.XX | X.XX | X.XX | X.XX | X.XX | XX |
| | VM1-Month 1 | XX | X.XX | X.XX | X.XX | X.XX | X.XX | XX |
| | V1-Month 3 | XX | X.XX | X.XX | X.XX | X.XX | X.XX | XX |
| | V2-Month 6 | XX | X.XX | X.XX | X.XX | X.XX | X.XX | XX |
| | V3-Month 9 | XX | X.XX | X.XX | X.XX | X.XX | X.XX | XX |
| | V4-Month 12 | XX | X.XX | X.XX | X.XX | X.XX | X.XX | XX |
| | V5-Month 15 | XX | X.XX | X.XX | X.XX | X.XX | X.XX | XX |
| | V6-Month 18 | XX | X.XX | X.XX | X.XX | X.XX | X.XX | XX |
| | V7-Month 21 | XX | X.XX | X.XX | X.XX | X.XX | X.XX | XX |
| | V8-Month 24 | XX | X.XX | X.XX | X.XX | X.XX | X.XX | XX |
| | V400- EOP-ind/con | XX | x.xx | X.XX | X.XX | X.XX | X.XX | XX |
| | V201-Month 27 * | XX | x.xx | X.XX | X.XX | X.XX | X.XX | XX |
| | V202-Month 30 * | XX | X.XX | X.XX | X.XX | X.XX | X.XX | XX |
| | V203-Month 33 * | XX | x.xx | X.XX | X.XX | X.XX | X.XX | XX |
| | V204-Month 36 * | XX | X.XX | X.XX | X.XX | X.XX | X.XX | XX |

<sup>-</sup> Unscheduled visits are taken into account. For each visit, the last available value is presented.

#### Programming note:

Repeat for ARM 1, ARM 2, Randomized Not Randomized

For: HDL (mmol/L), LDL (mmol/L), Glucose (mmol/L), Microalbumin (mg/L), HbA1c (%)

<sup>-</sup> Only visits corresponding to Induction/Consolidation phase are displayed.

<sup>-</sup> Perc.: Percentage.

<sup>\*</sup> For Arm 2 only.

Table 14.3-9.2.1 Total cholesterol shift table based on specific levels during Induction Consolidation – Full Analysis Set

| Analysis so | Baseline | | Worst post-baseline value | | | | |
|---|---|---|---|---|---|---|---|
| | | | Normal | | | | |
| | | n | cholesterolemia | | Hypercholesterolemia | | Missing |
| Treatment | | | n | (%) | n | (%) | n |
| Arm 1 | Normal cholesterolemia | xx | xx | (xx.x) | xx | (xx.x) | xx |
| (N=xxx) | Hypercholesterolemia | XX | XX | (xx.x) | XX | (xx.x) | XX |
| | Missing | XX | XX | (xx.x) | XX | (xx.x) | XX |
| | Total | XX | XX | (xx.x) | XX | (xx.x) | XX |
| Arm 2 | Normal cholesterolemia | XX | XX | (xx.x) | XX | (xx.x) | xx |
| (N=xxx) | Hypercholesterolemia | XX | XX | (xx.x) | XX | (xx.x) | XX |
| | Missing | XX | XX | (xx.x) | XX | (xx.x) | XX |
| | Total | XX | XX | (xx.x) | XX | (xx.x) | XX |
| Randomized (N=xxx) | Normal cholesterolemia | XX | XX | (xx.x) | XX | (xx.x) | xx |
| | Hypercholesterolemia | XX | XX | (xx.x) | XX | (xx.x) | XX |
| | Missing | XX | XX | (xx.x) | XX | (xx.x) | XX |
| | Total | XX | XX | (xx.x) | XX | (xx.x) | XX |
| Not Randomized | Normal cholesterolemia | XX | XX | (xx.x) | XX | (xx.x) | xx |
| (N=xxx) | Hypercholesterolemia | XX | XX | (xx.x) | XX | (xx.x) | XX |
| | Missing | XX | XX | (xx.x) | XX | (xx.x) | XX |
| | Total | XX | XX | (xx.x) | XX | (xx.x) | XX |
| Total | Normal cholesterolemia | XX | XX | (xx.x) | XX | (xx.x) | xx |
| (N=xxx) | Hypercholesterolemia | XX | XX | (xx.x) | XX | (xx.x) | XX |
| | Missing | XX | XX | (xx.x) | XX | (xx.x) | XX |
| | Total | XX | XX | (xx.x) | XX | (xx.x) | XX |

<sup>-</sup> Baseline is defined as the last available assessment before or at date of start of study treatment.

<sup>-</sup> Normal cholesterolemia defined as total cholesterol <=5.2 mmol/L; Hypercholesterolemia defined as total cholesterol >5.2 mmol/L.

<sup>-</sup> Percentage calculated by row, based on number of available patients at baseline and at least one non-missing post baseline value, (1-24 months for Arm 1, Not Randomized and Total, 1-36 months for Randomized and Arm 2).

<sup>&</sup>lt;< Programming note: use NTCHOBAS, NTCHOPSTin A LRS>>
## Table 14.3-9.2.2 Total cholesterol shift table based on specific levels during TFR phase — Subset of Full Analysis Set entering the TFR phase

<< Programming note: Same shell as table 14.3-9.2.1, for Arm 1, Arm 2 and Total, using NTCHOBAS2, NTCHOPST2 in A\_LRS and
footnotes:</pre>

- Baseline is defined as the last available assessment before or at date of start of study treatment.
- Normal cholesterolemia defined as total cholesterol <=5.2 mmol/L; Hypercholesterolemia defined as total cholesterol >5.2 mmol/L
- Percentage calculated by row, based on number of available patients at baseline and at least one non-missing post baseline value, (1-36 months for Arm 1, 1-24 months for Total and Arm 2).>>

## Table 14.3-9.2.3 Total cholesterol shift table based on specific levels during Re-treatment phase – Subset of Full Analysis Set entering the Re-treatment phase

<< Programming note: Same shell as table 14.3-9.2.1, for Arm 1, Arm 2 and Total, using NTCHOBAS3, NTCHOPST3 in A\_LRS and
footnotes:</pre>

- Baseline is defined as the last available assessment before or at date of start of study re-treatment.
- Normal cholesterolemia defined as total cholesterol <=5.2 mmol/L; Hypercholesterolemia defined as total cholesterol >5.2 mmol/L.
- Percentage calculated by row, based on number of available patients at baseline and at least one non-missing post baseline value, (1-36 months for Arm 1, 1-24 months for Total and Arm 2).>>

### Table 14.3-9.2.4 Total cholesterol shift table based on specific levels during TFR phase, SDV sensitivity – Subset of Full Analysis Set entering the TFR phase

<< Programming note: Same shell as Table 14.3-9.2.2, for SDV sensitivity analysis>>
Add footnote:

## Table 14.3-9.2.5 Total cholesterol shift table based on specific levels during Re-treatment phase, SDV sensitivity – Subset of Full Analysis Set entering the Re-treatment phase

<< Programming note: Same shell as Table 14.3-9.2.3, for SDV sensitivity analysis>> Add footnote:

Table 14.3-10.1.1 Fasting glucose shift table based on specific levels during Induction Consolidation – Full Analysis Set

| - | Baseli | ine | | Worst post-baseline value | | |
|---|---|---|---|---|---|---|
| Treatment | | n | Normal glycemia<br>n (%) | Hyperglycemia<br>n (%) | Diabetes<br>n (%) | Missing<br>n |
| Arm 1 | Normal glycemia | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX |
| (N=xxx) | Hyperglycemia | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX |
| | Diabetes | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX |
| | Missing | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX |
| | Total | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX |
| Arm 2 | Normal glycemia | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX |
| (N=xxx) | Hyperglycemia | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX |
| | Diabetes | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX |
| | Missing | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX |
| | Total | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX |
| Randomized | Normal glycemia | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX |
| (N=xxx) | Hyperglycemia | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx |
| | Diabetes | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx |
| | Missing | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx |
| | Total | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX |
| Not Randomized | Normal glycemia | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX |
| (N=xxx) | Hyperglycemia | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX |
| | Diabetes | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX |
| | Missing | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX |
| | Total | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX |
| Total | Normal glycemia | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX |
| (N=xxx) | Hyperglycemia | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX |
| | Diabetes | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX |
| | Missing | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX |
| | Total | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX |

<sup>-</sup> Baseline is defined as the last available assessment before or at date of start of study treatment.

<sup>-</sup> Normal glycemia defined as fasting glucose <5.6 mmol/L; Hyperglycemia defined as fasting glucose >=5.6-6.9 mmol/L; Diabetes defined as fasting glucose >6.9 mmol/L.

<sup>-</sup> Percentage calculated by row, based on number of available patients at baseline and at least one non-missing post baseline value, (1-24 months for Arm 1, Not Randomized and Total, 1-36 months for Arm 2).

<<Pre>rogramming note: use NGLUBAS and NGLUPST in A LRS >>

## Table 14.3-10.1.2 Fasting glucose shift table based on specific levels during TFR phase — Subset of Full Analysis Set entering the TFR phase

<< Programming note: Same shell as table 14.3-10.1.1, for Arm 1, Arm 2 and Total, using NGLUBAS2 and NGLUPST2 in A\_LRS and
footnotes:</pre>

- Baseline is defined as the last assessment in Ind/Cons phase
- Normal glycemia defined as fasting glucose <5.6 mmol/L; Hyperglycemia defined as fasting glucose >=5.6-6.9 mmol/L; Diabetes defined as fasting glucose >6.9 mmol/L.
- Percentage calculated by row, based on number of available patients at baseline and at least one. non-missing post baseline value, (1-24 months for Arm 1, 1-36 months for Total and Arm 2).>>

## Table 14.3-10.1.3 Fasting glucose shift table based on specific levels during Re-treatment phase — Subset of Full Analysis Set entering the Re-treatment phase

<< Programming note: Same shell as table 14.3-10.1.1, for Arm 1, Arm 2 and Total, using NGLUBAS3 and NGLUPST3 in A\_LRS and
footnotes:</pre>

- Baseline is defined as the last available assessment before or at date of start of study re-treatment. Normal glycemia defined as fasting glucose >= 5.6-6.9 mmol/L; Diabetes defined as fasting glucose > 6.9 mmol/L
- Percentage calculated by row, based on number of available patients at baseline and at least one non-missing post baseline value, (1-24 months for Arm 1, 1-36 months for Total and Arm 2).>>

## Table 14.3-10.1.4 Fasting glucose shift table based on specific levels during TFR phase, SDV sensitivity – Subset of Full Analysis Set entering the TFR phase

<< Programming note: Same shell as Table 14.3-10.1.2, for SDV sensitivity analysis>>
Add footnote:

## Table 14.3-10.1.5 Fasting glucose shift table based on specific levels during Re-treatment phase, SDV sensitivity – Subset of Full Analysis Set entering the Re-treatment phase

<< Programming note: Same shell as Table 14.3-10.1.3, for SDV sensitivity analysis>> Add footnote:

Table 14.3-11.1 Vital Signs during Induction Consolidation – Full Analysis Set

| Parameter | Visit | | Arm 1<br>N=xxx | Arm 2<br>N=xxx | Randomized<br>N=xxx | Not Randomized<br>N=xxx | Total<br>N=xxx |
|---|---|---|---|---|---|---|---|
| Body temperature (C) | Baseline | n<br>Missing<br>Mean<br>SD | xx<br>xx<br>xx.x | xx<br>xx<br>xx.x | xx<br>xx<br>xx.x | xx<br>xx<br>xx.x | xx<br>xx<br>xx.x |
| | | 25th Percentile<br>Median<br>75th Percentile<br>Min, Max | x.xx<br>xx.x<br>xx.x<br>xx.x<br>xx.x | x.xx<br>xx.x<br>xx.x<br>xx.x<br>xx.x | x.xx<br>xx.x<br>xx.x<br>xx.x<br>xx.x | x.xx<br>xx.x<br>xx.x<br>xx.x<br>xx.x | x.xx<br>xx.x<br>xx.x<br>xx.x<br>xx.x |
| | Month 3 | n<br> | xx | xx<br>··· | xx<br>··· | xx<br>··· | xx<br> |
| | • • • | | | | | | |
| | Month 24 | n<br>••• | xx<br>••• | xx<br>··· | xx<br>••• | xx<br> | xx<br>••• |
| | Month 27 | n<br>··· | Not applicable | xx<br> | xx<br> | Not applicable | xx<br>··· |
| | Month 30 | n | Not applicable | XX | XX | Not applicable | XX |
| | | • • • | | • • • | • • • | • • • | • • • |
| | Month 33 | n<br> | Not applicable | xx<br>··· | xx<br>··· | Not applicable | xx<br>··· |
| | Month 36 | n<br>••• | Not applicable | xx<br>··· | xx<br>••• | Not applicable | xx<br>··· |

| Novartis<br>RAP Module 7.1 | | | Confidential<br>6-May-2021 (14:35) | | | Protocol No CA | Page 317<br>MN107AIC0 |
|---|---|---|---|---|---|---|---|
| | Change from Baseline to Month 3 | n | xx | xx | xx | xx | xx |
| | | | ••• | | | • • • | |
| | Change from<br>Baseline to<br>Month 36 | n | Not applicable | xx | xx | Not applicable | xx |
| | | • • • | | • • • | • • • | | • • • |
| Sitting pulse (bpm) | Baseline | n | XX | XX | XX | XX | XX |
| | | • • • | ••• | • • • | • • • | • • • | • • • |
| Sitting blood<br>pressure Systolic<br>(mmHg) | Baseline | n | xx | xx | xx | xx | XX |
| | | • • • | ••• | • • • | • • • | • • • | • • • |
| | • • • | | | | | | |
| Sitting blood pressure Diastolic (mmHg) | Baseline | n | xx | xx | xx | xx | XX |
| | | • • • | • • • | • • • | | • • • | • • • |

<sup>-</sup> Baseline is defined as the last available assessment before or at date of start of study treatment

<sup>-</sup> Change from baseline: post baseline - baseline.

Novartis Confidential Page 318 RAP Module 7.1 Confidential Protocol No CAMN107AIC0

<< Programming note: use

Body Temperature: BTP1N (for PHASE=1), BASETP1N, CHGTP1N,

Sitting pulse: SPUNT1C (for PHASE=1), BASEPS1N, CHGPS1N

Sitting Diast BP: STNDBP1N (for PHASE=1), BASEDB1N, CHGDB1N

Sitting Syst BP: STNSBP1N (for PHASE=1), BASESB1N, CHGSB1N

from A\_VSN

For Missing use only records done(MRKEVL1C = 1 = Crossed) >>

#### Table 14.3-11.2 Vital Signs during TFR phase – Subset of Full Analysis Set entering the TFR phase

<< Same shell as table 14.3-11.1, for Arm 1, Arm 2 and Total, using

STNDBP1N (for PHASE=2), BASEDB2N, CHGDB2N

Body Temperature: BTP1N (for PHASE=2), BASETP2N, CHGTP2N,
Sitting pulse: SPUNT1C (for PHASE=2), BASEPS2N, CHGPS2N
Sitting Syst BP: STNSBP1N (for PHASE=2), BASESB2N, CHGSB2N

Sitting Diast BP: from A VSN

Change footnote to "Baseline is defined as the last treatment record in Ind/Cons phase">>

## Table 14.3-11.3 Vital Signs during Re-treatment phase – Subset of Full Analysis Set entering the Retreatment phase

<< Same shell as table 14.3-11.1, for Arm 1, Arm 2 and Total, using:

Body Temperature: BTP1N (for PHASE=3), BASETP3N, CHGTP3N,

Sitting pulse: SPUNT1C (for PHASE=3), BASEPS3N, CHGPS3N

Sitting Syst BP: STNSBP1N (for PHASE=3), BASESB3N, CHGSB3N

Sitting Diast BP: STNDBP1N (for PHASE=3), BASEDB3N, CHGDB3N

from A\_VSN

Change footnote to "Baseline is defined as the first treatment record during Re-treatment">>>

## Table 14.3-11.4 Vital Signs during TFR phase, SDV sensitivity – Subset of Full Analysis Set entering the TFR phase

<< Programming note: Same shell as Table 14.3-11.2, for SDV sensitivity analysis>>
Add footnote:

- SDV sensitivity: Excluding patient visits involved in SDV issues during final data review due to COVID-19.

## Table 14.3-11.5 Vital Signs during Re-treatment phase, SDV sensitivity – Subset of Full Analysis Set entering the Re-treatment phase

<< Programming note: Same shell as Table 14.3-11.3, for SDV sensitivity analysis>> Add footnote:

### Table 14.3-12.1 Survival follow-up – Full Analysis Set

| Visit | | Arm 1<br>N=xxx | Arm 2<br>N=xxx | Randomized<br>N=xxx | Not<br>Randomized | Total<br>N=xxx<br>n(%) |
|---|---|---|---|---|---|---|
| | | n (%) | n (%) | n (%) | N=xxx | |
| | | | | | n (%) | |
| FU-Month 3 | | N=xx | N=XX | N=xx | N=xx | N=xx |
| | Alive | | | | | |
| | Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Lost to follow-up | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Did patient undergo stem cell transplant? | | | | | |
| | Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Is the disease progressing to AP/BP ? | | | | | |
| | Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Is the patient receiving any TKI treatment ? | | | | | |
| | Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | If Yes | | | | | |
| | Nilotinib | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Imatinib | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Other | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| FU-Month 6 | | N=xx | N=xx | N=xx | N=xx | N=xx |
| | Patient alive | | | | | |

| Novartis RAP Module 7. | 1 | | Confidential<br>6-May-2021 (14:35) | | | | Page 322<br>Io CAMN107AIC0 |
|---|---|---|---|---|---|---|---|
| | | Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| • • • | | ••• | ••• | • • • | • • • | • • • | • • • |
| FU-Month 36 | | | | | | | |
| | Alive | | N=xx | N=xx | N=xx | N=xx | N=xx |
| | Yes | | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| • • • | | • • • | • • • | • • • | • • • | • • • | • • • |
| | | ••• | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

<sup>-</sup> Percentages calculated over available records for each FU visit.

#### Table 14.3-12.2 Survival follow-up, SDV sensitivity - Full Analysis Set

<< Programming note: Same shell as Table 14.3-12.1, for SDV sensitivity analysis>> Add footnote:

<sup>-</sup> SDV sensitivity: Excluding patient visits involved in SDV issues during final data review due to COVID-19.

### Table 14.3-13.1 Safety follow-up - Full analysis Set

| | Arm 1<br>N=xxx | Arm 2<br>N=xxx | Randomized<br>N=xxx | Not Randomized N=xxx | Total<br>N=xxx |
|---|---|---|---|---|---|
| Safety follow up perfomred? | n (%) | n (%) | n (%) | n (%) | n (%) |
| Yes, During Clinical visit | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Yes, During Telephone call | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| In case of Telephone call, Medical intervention necessary Yes No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

#### Table 14.3-13.2 Safety follow-up, SDV sensitivity - Full analysis Set

<< Programming note: Same shell as Table 14.3-13.1, for SDV sensitivity analysis>> Add footnote:

<sup>-</sup> SDV sensitivity: Excluding patient visits involved in SDV issues during final data review due to COVID-19.

#### Section 14.3.1 – Displays of adverse events

Figures (Section 14.3.1)

Figure 14.3.1-1.1 Kaplan-Meier analysis of time-to-first CVEs during the pre-randomization Induction/Consolidation phase – Full Analysis Set



<< Programming note: x-axis in Months, from 0 to 24 months >>

<< Programming note: 3 curves on the same plot: one for arm 1 patient and one for arm 2 patients, one for Not Randomized
patients>>

Add footnote:" - Presenting CVEs occurred within Pre-Randomization Ind/Cons phase only, excluding additional +30 days period used in TEAE outputs."

Figure 14.3.1-1.2 Kaplan-Meier analysis of time-to-first CVEs during the post-randomization consolidation phase (ARM 2) – Subset of Full Analysis Set randomized to Arm 2



<< Programming note: x-axis in Months, from 24 to 36 months >>

Add footnote: "- Presenting CVEs occurred within Post-Randomization consolidation phase only, excluding additional +30 days period used in TEAE outputs."

## Figure 14.3.1-1.3 Kaplan-Meier analysis of time-to-first CVEs during the the TFR phase – Subset of Full Analysis Set entering the TFR phase

<< Programming note:</pre>

The axis label should "Time since start of TFR phase (months)"

Months 0-36 for Arm 1, Months 0-24 for Arm 2

Split the curve into two: one for arm 1 patient and one for arm 2 patients >> Months 0-36 for Arm 1, Months 0-24 for Arm 2>>

## Figure 14.3.1-1.4 Kaplan-Meier analysis of time-to-first CVEs during the re-treatment phase – Subset of Full Analysis Set entering the re-treatment phase

<< Programming note: The axis label should "Time since start of Re-treatment phase (months)"

Months 0-36 for Arm 1, Months 0-24 for Arm 2

Split the curve into two: one for arm 1 patient and one for arm 2 patients >> Months 0-36 for Arm 1, Months 0-24 for Arm 2>> Add footnote: "- Presenting CVEs occurred within Re-treatment phase only, excluding additional +30 days period used in TEAE outputs."

Figure 14.3.1-2.1 Number of sorted events by HIS CD34+/CD38+ cells



Patients

#### Figure 14.3.1-2.2 Number of sorted events by PCR CD34+/CD38+ cells

<< Programming note: Same shell as Figure 14.3.1-2.1 replacing "HIS" by "PCR" >>

#### Figure 14.3.1-3.1 Number of sorted events by HIS CD34+/CD38- cells

<< Programming note: Same shell as Figure 14.3.1-2.1 replacing "CD34+/CD38+" by "CD34+/CD38-" >>

#### Figure 14.3.1-3.2 Number of sorted events by PCR CD34+/CD38- cells

<< Programming note: Same shell as Figure 14.3.1-2.2 replacing "CD34+/CD38+" by "CD34+/CD38-" >>

#### Figure 14.3.1-4.1 Number of sorted events by HIS Immunophenotypically aberrant CD34+ cells

<< Programming note: Same shell as Figure 14.3.1-2.1 replacing "CD34+/CD38+" by "Immunophenotypically aberrant CD34+" >>

#### Figure 14.3.1-4.2 Number of sorted events by PCR Immunophenotypically aberrant CD34+ cells

<< Programming note: Same shell as Figure 14.3.1-2.2 replacing "CD34+/CD38+" by "Immunophenotypically aberrant CD34+>>

#### Figure 14.3.1-5.1 Number of sorted events by HIS Immunophenotypically aberrant CD34- cells

<< Programming note: Same shell as Figure 14.3.1-2.1 replacing "CD34+/CD38+" by "Immunophenotypically aberrant CD34-" >>

#### Figure 14.3.1-5.2 Number of sorted events by PCR Immunophenotypically aberrant CD34- cells

<< Programming note: Same shell as Figure 14.3.1-2.2 replacing "CD34+/CD38+" by "Immunophenotypically aberrant CD34->>

Figure 14.3.1-6.1 Number of HIS+ subjects CD34+/CD38+ cells – LSC substudy Full Analysis Set



#### Figure 14.3.1-6.2 Number of PCR subjects CD34+/CD38+ cells – LSC substudy Full Analysis Set

<< Programming note: Same shell as Figure 14.3.1-6.1 replacing "HIS+" by "PCR" >>

#### Figure 14.3.1-7.1 Number of HIS+ subjects CD34+/CD38- cells – LSC substudy Full Analysis Set

<< Programming note: Same shell as Figure 14.3.1-6.1 replacing "CD34+/CD38+" by "CD34+/CD38-" >>

#### Figure 14.3.1-7.2 Number of PCR subjects CD34+/CD38- cells – LSC substudy Full Analysis Set

<< Programming note: Same shell as Figure 14.3.1-6.2 replacing "CD34+/CD38+" by "CD34+/CD38-" >>

## Figure 14.3.1-8.1 Number of HIS+ subjects Immunophenotypically aberrant CD34+ cells – LSC substudy Full Analysis Set

<< Programming note: Same shell as Figure 14.3.1-6.1 replacing "CD34+/CD38+" by "Immunophenotypically aberrant CD34+" >>

## Figure 14.3.1-8.2 Number of PCR subjects Immunophenotypically aberrant CD34+ cells – LSC substudy Full Analysis Set

<< Programming note: Same shell as Figure 14.3.1-6.2 replacing "CD34+/CD38+" by "Immunophenotypically aberrant CD34+" >>

## Figure 14.3.1-9.1 Number of HIS+ subjects Immunophenotypically aberrant CD34- cells – LSC substudy Full Analysis Set

<< Programming note: Same shell as Figure 14.3.1-6.1 replacing "CD34+/CD38+" by "Immunophenotypically aberrant CD34-" >>

### Figure 14.3.1-9.2 Number of PCR subjects Immunophenotypically aberrant CD34- cells – LSC substudy FAS

<< Programming note: Same shell as Figure 14.3.1-6.2 replacing "CD34+/CD38+" by "Immunophenotypically aberrant CD34-" >>

Figure 14.3.1-10 Number of patients with detectable LSC – LSC substudy Full Analysis Set



Detected cells by time point

#### Tables (Section 14.3.1)

Table 14.3.1-1.1 Overall summary of treatment-emergent adverse events occurring during pre-randomization Induction/consolidation phase – Full Analysis Set

| Adverse event category | Arm 1<br>N=xx | Arm 2<br>N=xx | Randomized<br>N=xx | Not Randomized<br>N=xx | Total<br>N=xx |
|---|---|---|---|---|---|
| Any adverse events | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any AE of special interest | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Grading of AEs NCI-CTCAE Grade 4 NCI-CTCAE Grade 3 NCI-CTCAE Grade 2 NCI-CTCAE Grade 1 NCI-CTCAE Missing | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) |
| Death | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AEs suspected to be related to nilotinib | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AEs leading to study drug discontinuation | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AEs requiring dosage adjustment or temporarily interruption | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Serious AEs | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Serious AEs suspected to be related to nilotinib | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Serious AEs leading to study drug discontinuation | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

<sup>-</sup> For patient # \_\_\_\_\_, due to reconciliation discrepancies, safety database reported AE term "Endometriosis" as a SAE, while in clinical database this AE was not recorded as an SAE.

Only TEAEs from pre-rand Ind./Cons. phase have been included in this table. A pat. with mult. occur. of an AE is counted only once in the AE category. Percentage based on the number of patients included in the analysis population (N). AESI CVEs (IHD), CVEs (PAOD), CVEs (ICD) and CVEs (others) are based on grouped MedDRA terms as described in the Case Retrieval Sheet. Treatment Arm 1/Arm 2: 24/36 months, Re-treatment max Arm 1/Arm 2: 36/24 months. Patient # reported as disc. Ind/Cons phase due to AE "Blast Crisis"- G2, should have been reported as disc. Ind/Cons phase due to Disease Progression, progression to Blast Crisis, as per Prot. For patient # AE "PHLEGMON FOOT - BIG TOE RIGHT" is reported as PT "Cellulitis" in the AE listing while it is reported as PT "Osteoarthritis" in the SAE listing. PT for the same AE has been wrongly decoded and reconciliation was not requiring a perfect match of the PT.

Table 14.3.1-1.2 Overall summary of treatment-emergent adverse events occurring during post-randomization consolidation phase (ARM 2) – Subset of Full Analysis Set randomized to Arm 2

| Adverse event category | N=xx |
|-------------------------------------------------------------|-----------|
| Any adverse events | xx (xx.x) |
| Any AE of special interest | xx (xx.x) |
| Grading of AEs | |
| NCI-CTCAE Grade 4 | xx (xx.x) |
| NCI-CTCAE Grade 3 | xx (xx.x) |
| NCI-CTCAE Grade 2 | xx (xx.x) |
| NCI-CTCAE Grade 1 | xx (xx.x) |
| NCI-CTCAE Missing | xx (xx.x) |
| Death | xx (xx.x) |
| AEs suspected to be related to nilotinib | xx (xx.x) |
| AEs leading to study drug discontinuation | xx (xx.x) |
| AEs requiring dosage adjustment or temporarily interruption | xx (xx.x) |
| Serious AEs | xx (xx.x) |
| Serious AEs suspected to be related to nilotinib | xx (xx.x) |
| Serious AEs leading to study drug discontinuation | xx (xx.x) |

<sup>-</sup> For patient # \_\_\_\_\_, due to reconciliation discrepancies, safety database reported AE term "Endometriosis" as a SAE, while in clinical database this AE was not recorded as an SAE.

<sup>-</sup> Only treatment emergent adverse events from post-randomization consolidation phase are included in this table.

<sup>-</sup> A patient with multiple occurrences of an AE is counted only once in the AE category.

<sup>-</sup> Percentage based on the number of patients included in the analysis population (N).

- AE of special interest CVEs (IHD), CVEs (PAOD), CVEs (ICD) and CVEs (others) are based on grouped MedDRA terms as described in the Case Retrieval Sheet. Patients randomized to Arm 2 have 12 months of treatment post-randomization and a maximum of 24 months of re-treatment. For patient AE "PHLEGMON FOOT - BIG TOE RIGHT" is reported as PT "Cellulitis" in the AE listing while it is reported as PT "Osteoarthritis" in the SAE listing. PT for the same AE has been wrongly decoded and reconciliation was not requiring a perfect match of the PT.

Table 14.3.1-1.3 Overall summary of treatment-emergent adverse events occurring during re-treatment phase – Subset of Full Analysis Set entering the re-treatment phase

| Adverse event category | Arm 1<br>N=xx | Arm 2<br>N=xx | Total<br>N=xx |
|---|---|---|---|
| | N-XX | N-XX | N-XX |
| Any adverse events | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any AE of special interest | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Grading of AEs | | | |
| NCI-CTCAE Grade 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| NCI-CTCAE Grade 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| NCI-CTCAE Grade 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| NCI-CTCAE Grade 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| NCI-CTCAE Missing | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Death | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AEs suspected to be related to nilotinib | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AEs leading to study drug discontinuation | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AEs requiring dosage adjustment or temporarily interruption | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Serious AEs | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Serious AEs suspected to be related to nilotinib | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Serious AEs leading to study drug discontinuation | xx (xx.x) | xx (xx.x) | xx (xx.x) |

<sup>-</sup> Only treatment emergent adverse events from re-treatment phase are included in this table.

<sup>-</sup> A patient with multiple occurrences of an AE is counted only once in the AE category.

<sup>-</sup> Percentage based on the number of patients included in the analysis population (N).

<sup>-</sup> Patients randomized to Arm 1 have 24 months of treatment and a maximum of 36 months of re-treatment.

<sup>-</sup> Patients randomized to Arm 2 have 36 months of treatment and a maximum of 24 months of re-treatment.

<sup>-</sup> AE of special interest CVEs (IHD), CVEs (PAOD), CVEs (ICD) and CVEs (others) are based on grouped MedDRA terms as described in the Case Retrieval Sheet.

Table 14.3.1-1.4 Overall summary of adverse events occurring during TFR phase – Subset of Full Analysis Set entering the TFR phase

| Adverse event category | Arm 1<br>N=xx | Arm 2<br>N=xx | Total<br>N=xx |
|---|---|---|---|
| Any adverse events | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any AE of special interest | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Grading of AEs | | | |
| NCI-CTCAE Grade 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| NCI-CTCAE Grade 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| NCI-CTCAE Grade 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| NCI-CTCAE Grade 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| NCI-CTCAE Missing | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Death | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AEs suspected to be related to nilotinib | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AE occurring within 30 days after TFR start <del>end</del> | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AE occurring after 30 days after TFR start end | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Serious AEs | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Serious AEs suspected to be related to nilotinib | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AE occurring within 30 days after TFR start | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AE occurring after 30 days after TFR start | xx (xx.x) | xx (xx.x) | xx (xx.x) |

<sup>-</sup> Only adverse events from TFR phase are included in this table.

<sup>-</sup> A patient with multiple occurrences of an AE is counted only once in the AE category.

<sup>-</sup> Percentage based on the number of patients included in the analysis population (N).

<sup>-</sup> Patients randomized to Arm 1 have 24 months of treatment and a maximum of 36 months of re-treatment.

<sup>-</sup> Patients randomized to Arm 2 have 36 months of treatment and a maximum of 24 months of re-treatment.

<sup>-</sup> AE of special interest CVEs (IHD), CVEs (PAOD), CVEs (ICD) and CVEs (others) are based on grouped MedDRA terms as described in the Case Retrieval Sheet.

#### Table 14.3.1-2.1 Overall summary of frequent [1] treatment-emergent adverse events occurring during prerandomization Induction/consolidation phase – Full Analysis Set

#### << Programming note: Same shell as table 14.3.1-1.1 adding the following footnote:</pre>

Only TEAEs from pre-rand Ind./Cons. phase have been included in this table. A pat. with mult. occur. of an AE is counted only once in the AE category. Perc. based on the number of pat. included in the analysis pop. (N).

AESI CVES (IHD), CVES (PAOD), CVES (ICD) and CVES (others) are based on grouped MedDRA terms as described in the CRS. Treatment Arm 1/Arm 2: 24/36 months, Re-treatment max Arm 1/Arm 2: 36/24 months. Patient # reported as disc. Ind/Cons phase due to AE "Blast Crisis"- G2, should have been reported as disc. Ind/Cons phase due to Disease Progression, progression to Blast Crisis, as per Prot. For patient # AE "PHLEGMON FOOT - BIG TOE RIGHT" is reported as PT "Cellulitis" in the AE listing while it is reported as PT "Osteoarthritis" in the SAE listing. PT for the same AE has been wrongly decoded and reconciliation was not requiring a perfect match of the PT.

[1] Frequent AE defined as an AE present at 5% or more for at least one treatment Arm.

#### Add following footnote at the end of last page:

- For patient # \_\_\_\_\_ due to reconciliation discrepancies, safety database reported AE term "Endometriosis" as a SAE, while in clinical database this AE was not recorded as an SAE.

## Table 14.3.1-2.2 Overall summary of frequent [1] treatment-emergent adverse events occurring during post-randomization consolidation phase (ARM 2) – Subset of Full Analysis Set randomized to Arm 2

<< Programming note: Same shell as table 14.3.1-1.2 adding the following footnote:
[1] Frequent AE defined as an AE present at 5% or more of the Arm2 patients.</pre>

## Table 14.3.1-2.3 Overall summary of frequent [1] treatment-emergent adverse events occurring during retreatment phase – Subset of Full Analysis Set entering the re-treatment phase

<< Programming note: Same shell as table 14.3.1-1.3 adding the following footnote:</pre>

[1] Frequent AE defined as an AE present at 5% or more for at least one treatment Arm.

## Table 14.3.1-2.4 Overall summary of frequent [1] adverse events occurring during TFR phase – Subset of Full Analysis Set entering the TFR phase

<< Programming note: Same shell as table 14.3.1-1.4 adding the following footnote:</pre>

[1] Frequent AE defined as an AE present at 5% or more for at least one treatment Arm.

Table 14.3.1-3.1.1 Treatment Emergent adverse events incidence, regardless of study drug relationship, occurring during pre-randomization Induction/consolidation phase by system organ class and preferred term - overall and maximum grade 3/4 – Full Analysis Set

| | Arr<br>N=2 | n 1<br>xxx | | m 2<br>xxx | | omized<br>xxx | | ndomized<br>xxx | Tot<br>N=> | |
|---|---|---|---|---|---|---|---|---|---|---|
| Primary system<br>organ class<br>Preferred term | All<br>grades<br>n (%) | Grade<br>3/4<br>n (%) | All<br>grades<br>n (%) | Grade<br>3/4<br>n (%) | All<br>grades<br>n (%) | Grade<br>3/4<br>n (%) | All<br>grades<br>n (%) | Grade<br>3/4<br>n (%) | All<br>grades<br>n (%) | Grade<br>3/4<br>n (%) |
| Any Primary<br>system organ<br>class | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Cardiac<br>disorders | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Angina pectoris | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Bradycardia NOS | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Oedema NOS | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Tachycardia NOS | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

<sup>-</sup> For patient # due to reconciliation discrepancies, safety database reported AE term "Endometriosis" as a SAE, while in clinical database this AE was not recorded as an SAE.

<sup>-</sup> Only TEAEs from pre-rand. Ind./Cons. phase have been included. Primary SOC are pres. alphab.; PTs are sorted within primary SOC in desc. freq. of 'All grades' column. Percentage based on the pop. number (N). Treatment Arm 1/Arm 2: 24/36 months, Re-trt max Arm 1/Arm 2: 36/24 months. A patient with mult. occur. of an AE is counted Only once in the AE cat.; A patient with mult. AEs within a primary SOC is counted only once in the total row. AEs occurring more than 30 days after last study trt exposure date are not summarized. Patient # reported as disc. Ind/Cons phase due to Disease Progression, progression to Blast Crisis, as per Prot. For patient # AE "PHLEGMON FOOT - BIG TOE RIGHT" is reported as PT "Cellulitis" in the AE listing while it is reported as PT "Osteoarthritis" in the SAE listing. PT for the same AE has been wrongly decoded and reconciliation was not requiring a perfect match of the PT.

## Table 14.3.1-3.1.2 Treatment Emergent adverse events occurrence, regardless of study drug relationship, occurring during pre-randomization Induction/consolidation phase by system organ class and preferred term - overall and maximum grade 3/4 – Full Analysis Set

<< Programming note: Same shell as table 14.3.1-3.1.1 but without percentages and use footnotes:</pre>

- Only treatment emergent adverse events from pre-rand. ind./cons. phase have been included in this table.
- Primary SOC are presented alphabetically; preferred terms are sorted within primary SOC in desc. frequency of 'All grades' column. Treatment Arm 1/Arm 2: 24/36 months, Re-trt max Arm 1/Arm 2: 36/24 months. AEs occurring more than 30 days after last study trt exposure date are not summarized.
- Patient # reported as disc. Ind/Cons phase due to AE "Blast Crisis" G2, should have been reported as disc. Ind/Cons phase due to Disease Progression, progression to Blast Crisis, as per Prot.
- For patient # AE "PHLEGMON FOOT BIG TOE RIGHT" is reported as PT "Cellulitis" in the AE listing while it is reported as PT "Osteoarthritis" in the SAE listing. PT for the same AE has been wrongly decoded and reconciliation was not requiring a perfect match of the PT.

#### Add following footnote at the end of last page:

- For patient # \_\_\_\_\_, due to reconciliation discrepancies, safety database reported AE term "Endometriosis" as a SAE, while in clinical database this AE was not recorded as an SAE.

Table 14.3.1-3.2.1 Treatment Emergent adverse events incidence, regardless of study drug relationship, occurring during post-randomization consolidation phase (ARM 2) by system organ class and preferred term - overall and maximum grade 3/4 – Subset of Full Analysis Set randomized to Arm 2

| | Arm | 1 2 |
|--------------------------------|-----------|-----------|
| | N=X | XXX |
| Primary system organ class | All | Grade |
| Preferred term | grades | 3/4 |
| | n (%) | n (%) |
| Any Primary system organ class | xx (xx.x) | xx (xx.x) |
| Cardiac disorders | xx (xx.x) | xx (xx.x) |
| Angina pectoris | xx (xx.x) | xx (xx.x) |
| Bradycardia NOS | xx (xx.x) | xx (xx.x) |
| Oedema NOS | xx (xx.x) | xx (xx.x) |
| Tachycardia NOS | xx (xx.x) | xx (xx.x) |

<sup>-</sup> Only treatment emergent adverse events from post-rand. cons. phase (ARM 2) are included in this table.

<sup>-</sup> Primary system organ classes are presented alphabetically; preferred terms are sorted within primary system organ class in descending frequency of 'All grades' column.

<sup>-</sup> Percentage based on the number of patients included in the analysis population (N).

<sup>-</sup> Treatment post-randomization Arm 2: 12 months, Re-treatment max Arm 2: 24 months.

<sup>-</sup> A patient with multiple occurrences of an AE is counted only once in the AE category.

<sup>-</sup> A patient with multiple adverse events within a primary system organ class is counted only once in the total row.

<sup>-</sup> Adverse events occurring more than 30 days after last study treatment exposure date are not summarized.

# Table 14.3.1-3.2.2 Treatment Emergent adverse events occurrence, regardless of study drug relationship, occurring during post-randomization consolidation phase (ARM 2) by system organ class and preferred term - overall and maximum grade 3/4 – Subset of Full Analysis Set randomized to Arm 2

<< Programming note: Same shell as table 14.3.1-3.2.1 but without percentages and use footnotes:

- Only treatment emergent adverse events from post-rand. cons. phase (ARM 2) are included in this table.
- Primary system organ classes are presented alphabetically; preferred terms are sorted within primary system organ class in descending frequency of 'All grades' column.
- Treatment post-randomization Arm 2: 12 months, Re-treatment max Arm 2: 24 months.
- Adverse events occurring more than 30 days after last study treatment exposure date are not summarized.

Table 14.3.1-3.3.1 Treatment-emergent adverse events incidence, regardless of study drug relationship, by system organ class and preferred term during re-treatment phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the re-treatment phase

| Primary system organ class<br>Preferred term | Arm 1<br>N=xx | | Arm 2<br>N=xx | | Total<br>N=xx | |
|---|---|---|---|---|---|---|
| | All grades<br>n (%) | Grade 3/4<br>n (%) | All grades<br>n (%) | Grade 3/4<br>n (%) | All grades<br>n (%) | Grade 3/4<br>n (%) |
| Any primary system organ class | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Cardiac disorders | | | | | | |
| Angina pectoris | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Bradycardia NOS | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Oedema NOS | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Tachycardia NOS | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| etc. | | | | | | |

<sup>-</sup> Only treatment emergent adverse events from re-treatment phase are included in this table.

<sup>-</sup> Primary system organ classes are alphabetically presented; preferred terms are sorted within primary system organ class in descending frequency of 'All grades' column.

<sup>-</sup> Percentage based on the number of patients included in the analysis population (N).

<sup>-</sup> Treatment Arm 1/Arm 2: 24/36 months, Re-treatment max Arm 1/Arm 2: 36/24 months.

<sup>-</sup> A patient with multiple occurrences of an AE is counted only once in the AE category.

<sup>-</sup> A patient with multiple AE within a primary system organ class is counted only once in the total row.

<sup>-</sup> Adverse events occurring more than 30 days after last study treatment exposure date are not summarized.

# Table 14.3.1-3.3.2 Treatment-emergent adverse events occurrence, regardless of study drug relationship, by system organ class and preferred term during re-treatment phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the re-treatment phase

<< Programming note: Same shell as table 14.3.1-3.3.1 but without percentages and use footnotes:</pre>

- Only treatment emergent adverse events from re-treatment phase are included in this table.
- Primary system organ classes are alphabetically presented; preferred terms are sorted within primary system organ class in descending frequency of 'All grades' column.
- Treatment Arm 1/Arm 2: 24/36 months, Re-treatment max Arm 1/Arm 2: 36/24 months.
- Adverse events occurring more than 30 days after last study treatment exposure date are not summarized.

## Table 14.3.1-3.4.1 Adverse events incidence, regardless of study drug relationship, by system organ class and preferred term during TFR phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the TFR phase

#### << Programming note: Same shell as table 14.3.1-3.3.1 and use footnote:</pre>

- Only adverse events from TFR phase are included in this table.
- Primary system organ classes are alphabetically presented; preferred terms are sorted within primary system organ class in descending frequency of 'All grades' column.
- Percentage based on the number of patients included in the analysis population (N).
- Treatment Arm 1/Arm 2: 24/36 months, Re-treatment max Arm 1/Arm 2: 36/24 months.
- A patient with multiple occurrences of an AE is counted only once in the AE category.
- A patient with multiple AE within a primary system organ class is counted only once in the total row.

## Table 14.3.1-3.4.2 Adverse events occurrence, regardless of study drug relationship, by system organ class and preferred term during TFR phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the TFR phase

<< Programming note: Same shell as table 14.3.1-3.4.3 but without percentages and use footnotes:</pre>

- Only adverse events from TFR phase are included in this table.
- Primary system organ classes are presented alphabetically; preferred terms are sorted within primary system organ class in descending frequency of 'All grades' column.
- Treatment Arm 1/Arm 2: 24/36 months, Re-treatment max Arm 1/Arm 2: 36/24 months.

# Table 14.3.1-3.5.1 Frequent [1] Treatment Emergent adverse events incidence, regardless of study drug relationship occurring during pre-randomization Induction/consolidation phase by system organ class and preferred term - overall and maximum grade 3/4 – Full Analysis Set

<< Programming note: Same shell as table 14.3.1-3.1.1 >>

Only TEAEs from pre-rand Ind./Cons. phase have been included in this table. A pat. with mult. occur. of an AE is counted only once in the AE category. Perc. based on the number of pat. included in the analysis pop. (N).

AESI CVES (IHD), CVES (PAOD), CVES (ICD) and CVES (others) are based on grouped MedDRA terms as described in the CRS. Treatment Arm 1/Arm 2: 24/36 months, Re-treatment max Arm 1/Arm 2: 36/24 months.

Patient # Parameter are provided as disc. Ind/Cons phase due to AE "Blast Crisis" - G2, should have been reported as disc.

Ind/Cons phase due to Disease Progression, progression to Blast Crisis, as per Prot. For patient AE "PHLEGMON FOOT - BIG TOE RIGHT" is reported as PT "Cellulitis" in the AE listing while it is reported as PT "Osteoarthritis" in the SAE listing. PT for the same AE has been wrongly decoded and reconciliation was not requiring a perfect match of the PT.

[1] Frequent AE defined as an AE present at 5% or more for at least one treatment Arm.

Programming Note: Consider only AEs with >5% for Total group at the level of Preferred Term.

Re-calculate Primay SOC and Any Primary SOC frequencies accordingly, based on the selected AEs only.

Table 14.3.1-3.5.2 Frequent [1] Treatment Emergent adverse events incidence, regardless of study drug relationship occurring during post-randomization consolidation phase (ARM 2) by system organ class and preferred term- overall and maximum grade 3/4 – Subset of Full Analysis Set randomized to Arm 2

<< Programming note: Same shell as table 14.3.1-3.2.1 adding the following footnote:
[1] Frequent AE defined as an AE present at 5% or more of the Arm2 patients.</pre>

Programming Note: Consider only AEs with >5% for Total group at the level of Preferred Term.

Re-calculate Primay SOC and Any Primary SOC frequencies accordingly, based on the selected AEs only.
## Table 14.3.1-3.5.3 Frequent [1] Treatment Emergent adverse events incidence, regardless of study drug relationship occurring during re-treatment phase by system organ class and preferred term- overall and maximum grade 3/4 – Subset of Full Analysis Set entering the re-treatment phase

<< Programming note: Same shell as table 14.3.1-3.3.1 adding the following footnote:
[1] Frequent AE defined as an AE present at 5% or more for at least one treatment Arm.
Programming Note: Consider only AEs with >5% for Total group at the level of Preferred Term.
Re-calculate Primay SOC and Any Primary SOC frequencies accordingly, based on the selected AEs only.

## Table 14.3.1-3.5.4 Frequent [1] adverse events incidence, regardless of study drug relationship occurring during TFR phase by system organ class and preferred term - overall and maximum grade 3/4 – Subset of Full Analysis Set entering the TFR phase

<< Programming note: Same shell as table 14.3.1-3.4.1 adding the following footnote:
[1] Frequent AE defined as an AE present at 5% or more for at least one treatment Arm.
Programming Note: Consider only AEs with >5% for Total group at the level of Preferred Term.
Re-calculate Primay SOC and Any Primary SOC frequencies accordingly, based on the selected AEs only.

## Table 14.3.1-4.1.1 Serious treatment-emergent adverse events incidence, regardless of study drug relationship, by system organ class and preferred term during pre-randomization Induction/consolidation phase – overall and maximum grade 3/4 –Full Analysis Set

#### Add following footnote at the end of last page:

- For patient # \_\_\_\_\_, due to reconciliation discrepancies, safety database reported AE term "Endometriosis" as a SAE, while in clinical database this AE was not recorded as an SAE.

## Table 14.3.1-4.1.2 Serious treatment-emergent adverse events occurence, regardless of study drug relationship, by system organ class and preferred term during pre-randomization Induction/consolidation phase – overall and maximum grade 3/4 –Full Analysis Set

<< Programming note: Same shell as table 14.3.1-3.1.2 >>

- Only TEAEs from pre-rand. ind./cons. phase have been included in this table. Prim. SOC are pres. alphabetically; preferred terms are sorted within primary system organ class in descending frequency of 'All grades' column.
- Treatment Arm 1/Arm 2: 24/36 months, treatment free remission max Arm 1/Arm 2: 36/24 months.
- Adverse events occurring more than 30 days after last study treatment exposure date are not summarized.

  Patient # reported as disc. Ind/Cons phase due to AE "Blast Crisis" G2, should have been reported as disc. Ind/Cons phase due to Disease Progression, progr. to Blast Crisis, as per Prot. For patient # AE "PHLEGMON FOOT BIG TOE RIGHT" is reported as PT "Cellulitis" in the AE listing while it is reported as PT "Osteoarthritis" in the SAE listing. PT for the same AE has been wrongly decoded and reconciliation was not requiring a perfect match of the PT.

#### Add following footnote at the end of last page:

- For patient \_\_\_\_\_, due to reconciliation discrepancies, safety database reported AE term "Endometriosis" as a SAE, while in clinical database this AE was not recorded as an SAE.

Table 14.3.1-4.2.1 Serious treatment-emergent adverse events incidence, regardless of study drug relationship, by system organ class and preferred term during post-randomization consolidation phase (ARM 2) – overall and maximum grade 3/4 – Subset of Full Analysis Set randomized to Arm 2

<< Programming note: Same shell as table 14.3.1-3.2.1>>

Table 14.3.1-4.2.2 Serious treatment-emergent adverse events occurrence, regardless of study drug relationship, by system organ class and preferred term during post-randomization consolidation phase (ARM 2) – overall and maximum grade 3/4 – Subset of Full Analysis Set randomized to Arm 2

<< Programming note: Same shell as table 14.3.1-3.2.2 >>

Table 14.3.1-4.3.1 Serious treatment-emergent adverse events incidence, regardless of study drug relationship, by system organ class and preferred term during re-treatment phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the re-treatment phase

<< Programming note: Same shell as table 14.3.1-3.3.1 >>

Table 14.3.1-4.3.2 Serious treatment-emergent adverse events occurrence, regardless of study drug relationship, by system organ class and preferred term during re-treatment phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the re-treatment phase

<< Programming note: Same shell as table 14.3.1-3.3.2 >>

Table 14.3.1-4.4.1 Serious adverse events incidence, regardless of study drug relationship, by system organ class and preferred term during TFR phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the TFR phase

<< Programming note: Same shell as table 14.3.1-3.4.1>>

Table 14.3.1-4.4.2 Serious adverse events occurence, regardless of study drug relationship, by system organ class and preferred term during TFR phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the TFR phase

<< Programming note: Same shell as table 14.3.1-3.4.2>>

Table 14.3.1-4.5.1 Frequent [1] Serious Treatment Emergent adverse events incidence, regardless of study drug relationship occurring during pre-randomization Induction/consolidation phase by system organ class and preferred term - overall and maximum grade 3/4 – Full Analysis Set

<< Programming note: Same shell as table 14.3.1-3.5.1>>
Programming Note: Consider only AEs with >5% for one or more treatment Arms at the level of Preferred Term.
Re-calculate Primay SOC and Any Primary SOC frequencies accordingly, based on the selected AEs only.

Table 14.3.1-4.5.2 Frequent [1] Serious Treatment Emergent adverse events incidence, regardless of study drug relationship occurring during post-randomization consolidation phase (ARM 2) by system organ class and preferred term - overall and maximum grade 3/4 – Subset of Full Analysis Set randomized to Arm 2

<< Programming note: Same shell as table 14.3.1-3.5.2>>
Programming Note: Consider only AEs with >5% for or more treatment Arms at the level of Preferred Term.
Re-calculate Primay SOC and Any Primary SOC frequencies accordingly, based on the selected AEs only.

Table 14.3.1-4.5.3 Frequent [1] Serious Treatment Emergent adverse events incidence, regardless of study drug relationship occurring during re-treatment phase by system organ class and preferred term - overall and maximum grade 3/4 — Subset of Full Analysis Set entering the re-treatment phase

<< Programming note: Same shell as table 14.3.1-3.5.3 >>
Programming Note: Consider only AEs with >5% for or more treatment Arms at the level of Preferred Term.
Re-calculate Primay SOC and Any Primary SOC frequencies accordingly, based on the selected AEs only.

Table 14.3.1-4.5.4 Frequent [1] Serious adverse events incidence, regardless of study drug relationship occurring during TFR phase by system organ class and preferred term - overall and maximum grade 3/4 – Subset of Full Analysis Set entering the TFR phase

<< Programming note: Same shell as table 14.3.1-3.5.4 >>
Programming Note: Consider only AEs with >5% for or more treatment Arms at the level of Preferred Term.
Re-calculate Primay SOC and Any Primary SOC frequencies accordingly, based on the selected AEs only.

## Table 14.3.1-4.6.1 Serious treatment-emergent adverse events incidence, suspected to be study drug related, by system organ class and preferred term during pre-randomization Induction/consolidation phase – overall and maximum grade 3/4 –Full Analysis Set

<< Programming note: Same shell as table 14.3.1-3.1.1 >>

- Only TEAEs from pre-rand. Ind./Cons. phase have been included. Primary SOC are pres. alphab.; PTs are sorted within primary SOC in desc. freq. of 'All grades' column. Percentage based on the pop. number (N). Treatment Arm 1/Arm 2: 24/36 months, Re-trt max Arm 1/Arm 2: 36/24 months. A patient with mult. occur. of an AE is counted Only once in the AE cat.; A patient with mult. AEs within a primary SOC is counted only once in the total row. AEs occurring more than 30 days after last study trt exposure date are not summarized. Patient # reported as disc. Ind/Cons phase due to AE "Blast Crisis" - G2, should have been reported as disc. Ind/Cons phase due to Disease Progression, progression to Blast Crisis, as per Prot. For patient # AE "PHLEGMON FOOT - BIG TOE RIGHT" is reported as PT "Cellulitis" in the AE listing while it is reported as PT "Osteoarthritis" in the SAE listing. PT for the same AE has been wrongly decoded and reconciliation was not requiring a perfect match of the PT.

#### Add following footnote at the end of last page:

- For patient , due to reconciliation discrepancies, safety database reported AE term "Endometriosis" as a SAE, while in clinical database this AE was not recorded as an SAE.

## Table 14.3.1-4.6.2 Serious treatment-emergent adverse events occurence, suspected to be study drug related, by system organ class and preferred term during pre-randomization Induction/consolidation phase – overall and maximum grade 3/4 –Full Analysis Set

<< Programming note: Same shell as table 14.3.1-3.1.2 >>

- Only TEAEs from post-randomization consolidation phase are included in this table. A patient with multiple occurrences of an AE is counted only once in the AE category. Percentage based on the number of patients included in the analysis population (N). AE of special interest CVEs (IHD), CVEs (PAOD), CVEs (ICD) and CVEs (others) are based on grouped MedDRA terms as described in the Case Retrieval Sheet. Patients randomized to Arm 2 have 12 months of treatment post-randomization and a maximum of 24 months of re-treatment. Patient # reported as disc.

Ind/Cons phase due to AE "Blast Crisis" - G2, should have been reported as disc. Ind/Cons phase due to Disease Progression, progression to Blast Crisis, as per Prot. For patient # AE "PHLEGMON FOOT - BIG TOE RIGHT" is reported as PT "Cellulitis" in the AE listing while it is reported as PT "Osteoarthritis" in the SAE listing.

PT for the same AE has been wrongly decoded and reconciliation was not requiring a perfect match of the PT.

#### Add following footnote at the end of last page:

- For patient due to reconciliation discrepancies, safety database reported AE term "Endometriosis" as a SAE, while in clinical database this AE was not recorded as an SAE.

Table 14.3.1-4.7.1 Serious treatment-emergent adverse events incidence, suspected to be study drug related, by system organ class and preferred term during post-randomization consolidation phase (ARM 2) – overall and maximum grade 3/4 – Subset of Full Analysis Set randomized to Arm 2

<< Programming note: Same shell as table 14.3.1-3.2.1 >>

Table 14.3.1-4.7.2 Serious treatment-emergent adverse events occurrence, suspected to be study drug related, by system organ class and preferred term during post-randomization consolidation phase (ARM 2) – overall and maximum grade 3/4 – Subset of Full Analysis Set randomized to Arm 2

<< Programming note: Same shell as table 14.3.1-3.2.2 >>

Table 14.3.1-4.8.1 Serious treatment-emergent adverse events incidence, suspected to be study drug related, by system organ class and preferred term during re-treatment phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the re-treatment phase

<< Programming note: Same shell as table 14.3.1-3.3.1 >>

Table 14.3.1-4.8.2 Serious treatment-emergent adverse events occurrence, suspected to be study drug related, by system organ class and preferred term during re-treatment phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the re-treatment phase

<< Programming note: Same shell as table 14.3.1-3.3.2>>

Table 14.3.1-4.9.1 Serious adverse events incidence, suspected to be study drug related, by system organ class and preferred term during TFR phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the TFR phase

<< Programming note: Same shell as table 14.3.1-3.4.1 >>

## Table 14.3.1-4.9.2 Serious adverse events occurrence, suspected to be study drug related, by system organ class and preferred term during TFR phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the TFR phase

<< Programming note: Same shell as table 14.3.1-3.4.2>>

## Table 14.3.1-5.1.1 Treatment-emergent adverse events incidence leading to study drug discontinuation by system organ class and preferred term during pre-randomization Induction/Consolidation phase – overall and maximum grade 3/4 –Full Analysis Set

#### << Programming note: Same shell as table 14.3.1-3.1.1>>

- Only TEAEs from pre-rand. ind./cons. phase have been included in this table. Primary SOC are presented alphabetically; PTs are sorted within primary SOC in descending frequency of 'All grades' column.
- Percentage based on the number of patients included in the analysis population (N).
- Treatment Arm 1/Arm 2: 24/36 months, Re-treatment max Arm 1/Arm 2: 36/24 months.
- A patient with multiple occurrences of an AE is counted only once in the AE category.
- A patient with multiple AEs within a primary system organ class is counted only once in the total row
- Adverse events occurring more than 30 days after last study treatment exposure date are not summarized.
- Patient reported as disc. Ind/Cons phase due to AE "Blast Crisis" G2, should have been reported as disc. Ind/Cons phase due to Disease Progression, progression to Blast Crisis, as per Prot.

#### Add following footnote at the end of last page:

- For patient # \_\_\_\_\_, due to reconciliation discrepancies, safety database reported AE term "Endometriosis" as a SAE, while in clinical database this AE was not recorded as an SAE.

## Table 14.3.1-5.1.2 Treatment-emergent adverse events occurence leading to study drug discontinuation by system organ class and preferred term during pre-randomization Induction/Consolidation phase – overall and maximum grade 3/4 –Full Analysis Set

<< Programming note: Same shell as table 14.3.1-3.1.2>>

- Only treatment emergent adverse events from pre-rand. ind./cons. phase have been included in this table.
- Primary system organ classes are presented alphabetically; preferred terms are sorted within primary system organ class in descending frequency of 'All grades' column.
- Treatment Arm 1/Arm 2: 24/36 months, Re-treatment max Arm 1/Arm 2: 36/24 months.
- Adverse events occurring more than 30 days after last study treatment exposure date are not summarized.
- Patient # reported as disc. Ind/Cons phase due to AE "Blast Crisis" G2, should have been reported as disc. Ind/Cons phase due to Disease Progression, progression to Blast Crisis, as per Prot.

#### Add following footnote at the end of last page:

- For patient # \_\_\_\_\_, due to reconciliation discrepancies, safety database reported AE term "Endometriosis" as a SAE, while in clinical database this AE was not recorded as an SAE.

Table 14.3.1-5.2.1 Treatment-emergent adverse events incidence leading to study drug discontinuation by system organ class and preferred term during post-randomization phase (ARM 2) – overall and maximum grade 3/4 – Subset of Full Analysis Set randomized to Arm 2

<< Programming note: Same shell as table 14.3.1-3.2.1 >>

Table 14.3.1-5.2.2 Treatment-emergent adverse events occurrence leading to study drug discontinuation by system organ class and preferred term during post-randomization phase (ARM 2)— overall and maximum grade 3/4 – Subset of Full Analysis Set randomized to Arm 2

<< Programming note: Same shell as table 14.3.1-3.2.2 >>

Table 14.3.1-5.3.1 Treatment-emergent adverse events incidence leading to study drug discontinuation by system organ class and preferred term during re-treatment phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the re-treatment phase

<< Programming note: Same shell as table 14.3.1-3.3.1 >>

Table 14.3.1-5.3.2 Treatment-emergent adverse events occurrence leading to study drug discontinuation by system organ class and preferred term during re-treatment phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the re-treatment phase

<< Programming note: Same shell as table 14.3.1-3.3.2 >>

Table 14.3.1-6.1.1 Treatment-emergent adverse events incidence requiring dosage adjustment or temporarily interruption by system organ class and preferred term during pre-randomization Induction/consolidation phase – overall and maximum grade 3/4 –Full Analysis Set

<< Programming note: Same shell as table 14.3.1-3.1.1 >>

- Only TEAEs from pre-rand. Ind./Cons. phase have been included. Primary SOC are pres. alphab.; PTs are sorted within primary SOC in desc. freq. of 'All grades' column. Percentage based on the pop. number (N). Treatment Arm 1/Arm 2: 24/36 months, Re-trt max Arm 1/Arm 2: 36/24 months. A patient with mult. occur. of an AE is counted Only once in the AE cat.; A patient with mult. AEs within a primary SOC is counted only once in the total row. AEs occurring more than 30 days after last study trt exposure date are not summarized. Patient # reported as disc. Ind/Cons phase due to AE "Blast Crisis" - G2, should have been reported as disc. Ind/Cons phase due to Disease Progression, progression to Blast Crisis, as per Prot. For patient # AE "PHLEGMON FOOT - BIG TOE RIGHT" is reported as PT "Cellulitis" in the AE listing while it is reported as PT "Osteoarthritis" in the SAE listing. PT for the same AE has been wrongly decoded and reconciliation was not requiring a perfect match of the PT.

Add following footnote at the end of last page:

- For patient # \_\_\_\_\_, due to reconciliation discrepancies, safety database reported AE term "Endometriosis" as a SAE, while in clinical database this AE was not recorded as an SAE.

## Table 14.3.1-6.1.2 Treatment-emergent adverse events occurrence requiring dosage adjustment or temporarily interruption by system organ class and preferred term during pre-randomization Induction/consolidation phase – overall and maximum grade 3/4 –Full Analysis Set

<< Programming note: Same shell as table 14.3.1-3.1.2 >>

- Only treatment emergent adverse events from pre-rand. ind./cons. phase have been included in this table.
- Primary SOC are presented alphabetically; preferred terms are sorted within primary SOC in desc. frequency of 'All grades' column. Treatment Arm 1/Arm 2: 24/36 months, Re-trt max Arm 1/Arm 2: 36/24 months. AEs occurring more than 30 days after last study trt exposure date are not summarized.
- Patient # \_\_\_\_\_ reported as disc. Ind/Cons phase due to AE "Blast Crisis"- G2, should have been reported as disc. Ind/Cons phase due to Disease Progression, progression to Blast Crisis, as per Prot.
- For patient # AE "PHLEGMON FOOT BIG TOE RIGHT" is reported as PT "Cellulitis" in the AE listing while it is reported as PT "Osteoarthritis" in the SAE listing. PT for the same AE has been wrongly decoded and reconciliation was not requiring a perfect match of the PT.

#### Add following footnote at the end of last page:

- For patient # \_\_\_\_\_, due to reconciliation discrepancies, safety database reported AE term "Endometriosis" as a SAE, while in clinical database this AE was not recorded as an SAE.

Table 14.3.1-6.2.1 Treatment-emergent adverse events incidence requiring dosage adjustment or temporarily interruption by system organ class and preferred term during post-randomization consolidation phase (ARM 2) – overall and maximum grade 3/4 – Subset of Full Analysis Set randomized to Arm 2

<- Programming note: Same shell as table 14.3.1-3.2.1 >>

Table 14.3.1-6.2.2 Treatment-emergent adverse events occurrence requiring dosage adjustment or temporarily interruption by system organ class and preferred term during post-randomization consolidation phase (ARM 2) – overall and maximum grade 3/4 – Subset of Full Analysis Set randomized to Arm 2

<< Programming note: Same shell as table 14.3.1-3.2.2>>

Table 14.3.1-6.3.1 Treatment-emergent adverse events incidence requiring dosage adjustment or temporarily interruption by system organ class and preferred term during re-treatment phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the re-treatment phase

<< Programming note: Same shell as table 14.3.1-3.3.1 >>

Table 14.3.1-6.3.2 Treatment-emergent adverse events occurrence requiring dosage adjustment or temporarily interruption by system organ class and preferred term during re-treatment phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the re-treatment phase

<< Programming note: Same shell as table 14.3.1-3.3.2 >>

Table 14.3.1-6.4.1 Treatment-emergent adverse events of interest incidence, regardless of study drug relationship, by specific group and preferred term during Pre-randomization Induction/consolidation phase –by treatment arm, overall and maximum grade 3/4 – Full Analysis Set

| | | m 1<br>xxx | | m 2<br>xxx | | omized<br>xxx | | ndomized<br>xxx | | tal<br>xxx |
|---|---|---|---|---|---|---|---|---|---|---|
| Specific group<br>Preferred term | All<br>grades<br>n (%) | Grade<br>3/4<br>n (%) | All<br>grades<br>n (%) | Grade<br>3/4<br>n (%) | All<br>grades<br>n (%) | Grade<br>3/4<br>n (%) | All<br>grades<br>n (%) | Grade<br>3/4<br>n (%) | All<br>grades<br>n (%) | Grade<br>3/4<br>n (%) |
| All AESI | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Group 1 | | | | | | | | | | |
| PT1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Group 2 | | | | | | | | | | |
| PT1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT2<br> | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

<sup>-</sup> Only treatment emergent adverse events from pre-rand. ind./cons. phase have been included in this table.

<< Programming note: The below groups of AEs of special interest will be displayed:

<sup>-</sup> Specific groupings are presented alphabetically; preferred terms are sorted within each group in descending frequency of 'All grades' column. Percentage based on the number of patients included in the analysis population (N).

<sup>-</sup> Treatment Arm 1/Arm 2: 24/36 months, Re-treatment max Arm 1/Arm 2: 36/24 months.

<sup>-</sup> A patient with multiple occurrences of an AE is counted only once in the AE category. A patient with multiple adverse events within a group is counted only once in the total row. AE of special interest CVEs (IHD), CVEs (PAOD), CVEs (ICD) and CVEs (others) are based on grouped MedDRA terms as described in the Case Retrieval Sheet. AEs occurring more than 30 days after last study treatment exposure date are not summarized.

<sup>-</sup>CVEs (IHD: Ischemic heart disease)

<sup>-</sup>CVEs (PAOD: Peripheral arterial occlusive disease)

<sup>-</sup>CVEs (ICE: Ischemic cerebrovascular events)

<sup>-</sup>CVEs (Others)

## Table 14.3.1-6.4.2 Treatment-emergent adverse events of interest occurrence, regardless of study drug relationship, by specific group and preferred term during Pre-randomization Induction/consolidation phase – by treatment arm, overall and maximum grade 3/4 –Full Analysis Set

<< Programming note: Same shell as table 14.3.1-6.4.1 but without percentages, use footnotes:</pre>

- Only treatment emergent adverse events from pre-rand. ind./cons. phase have been included in this table.
- Specific groupings are presented alphabetically; preferred terms are sorted within each group in descending frequency of 'All grades' column.
- Treatment Arm 1/Arm 2: 24/36 months, Re-treatment max Arm 1/Arm 2: 36/24 months.
- AE of special interest CVEs (IHD), CVEs (PAOD), CVEs (ICD) and CVEs (others) are based on grouped MedDRA terms as described in the Case Retrieval Sheet. AEs occurring more than 30 days after last study treatment exposure date are not summarized.

Table 14.3.1-6.5.1 Treatment-emergent adverse events of interest incidence by specific group and preferred term during post-randomization consolidation phase (ARM 2) – overall and maximum grade 3/4 – Subset of Full Analysis Set randomized to Arm 2

| Specific group Preferred term | Arm 2 | |
|-------------------------------|------------|-----------|
| | 1 | √=xx |
| | All grades | Grade 3/4 |
| | n (%) | n (%) |
| All AESI | xx (xx.x) | xx (xx.x) |
| Group 1 | | |
| PT 1 | xx (xx.x) | xx (xx.x) |
| PT 2 | xx (xx.x) | xx (xx.x) |
| ect | xx (xx.x) | xx (xx.x) |
| Group 2 | | |
| PT 1 | xx (xx.x) | xx (xx.x) |
| PT 2 | xx (xx.x) | xx (xx.x) |
| ect | xx (xx.x) | xx (xx.x) |
| ect | | |

<sup>-</sup> Only treatment emergent adverse events from post-rand. cons. phase are included in this table.

<sup>-</sup> Specific groups are alphabetically presented; preferred terms are sorted within each group in descending frequency of 'All grades' column. Percentage based on the number of patients included in the analysis population (N).

<sup>-</sup> Treatment post-randomization Arm 2: 12 months, Re-treatment max Arm 2: 24 months.

<sup>-</sup> A patient with multiple occurrences of an AE is counted only once in the AE category. A patient with multiple adverse events within a group is counted only once in the total row. AE of special interest CVEs (IHD), CVEs (PAOD), CVEs (ICD) and CVEs (others) are based on grouped MedDRA terms as described in the Case Retrieval Sheet. AEs occurring more than 30 days after last study treatment exposure date are not summarized.

## Table 14.3.1-6.5.2 Treatment-emergent adverse events of interest occurrence, by specific group and preferred term during post-randomization consolidation phase (ARM 2) – overall and maximum grade 3/4 – Subset of Full Analysis Set randomized to Arm 2

<< Programming note: Same shell as table 14.3.1-6.5.1 but without percentages, use footnotes:</pre>

- Only treatment emergent adverse events from post-rand. cons. phase are included in this table.
- Specific groups are alphabetically presented; preferred terms are sorted within each group in descending frequency of 'All grades' column.
- Treatment post-randomization Arm 2: 12 months, Re-treatment max Arm 2: 24 months. AE of special interest CVEs (IHD), CVEs (PAOD), CVEs (ICD) and CVEs (others) are based on grouped MedDRA terms as described in the Case Retrieval Sheet.
- AEs occurring more than 30 days after last study treatment exposure date are not summarized.

Table 14.3.1-6.6.1 Treatment-emergent adverse events of interest incidence by specific group and preferred term during re-treatment phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the re-treatment phase

| Specific group Preferred term | | m 1<br>=xx | Arm<br>N=: | | Total<br>N=xx | |
|---|---|---|---|---|---|---|
| | All grades | Grade 3/4 | All grades | Grade 3/4 | All grades | Grade 3/4 |
| | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| All AESI | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Group 1 | | | | | | |
| PT 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ect | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Group 2 | | | | | | |
| PT 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ect | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ect | | | | | | |

<sup>-</sup> Only treatment emergent adverse events from re-treatment phase are included in this table.

<sup>-</sup> Specific groups are alphabetically presented; preferred terms are sorted within each group in descending frequency of 'All grades' column. Percentage based on the number of patients included in the analysis population (N).

<sup>-</sup> Treatment Arm 1/Arm 2: 24/36 months, Re-treatment max Arm 1/Arm 2: 36/24 months.

<sup>-</sup> A patient with multiple occurrences of an AE is counted only once in the AE category. A patient with multiple adverse events within a group is counted only once in the total row. AE of special interest CVEs (IHD), CVEs (PAOD), CVEs (ICD) and CVEs (others) are based on grouped MedDRA terms as described in the Case Retrieval Sheet.AEs occurring more than 30 days after last study treatment exposure date are not summarized.

## Table 14.3.1-6.6.2 Treatment-emergent adverse events of interest occurrence by specific group and preferred term during re-treatment phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the re-treatment phase

<< Programming note: Same shell as table 14.3.1-6.6.1 but without percentages, use footnotes:</pre>

- Only treatment emergent adverse events from re-treatment phase are included in this table.
- Specific groups are alphabetically presented; preferred terms are sorted within each group in descending frequency of 'All grades' column.
- Treatment Arm 1/Arm 2: 24/36 months, Re-treatment max Arm 1/Arm 2: 36/24 months.
- AE of special interest CVEs (IHD), CVEs (PAOD), CVEs (ICD) and CVEs (others) are based on grouped MedDRA terms as described in the Case Retrieval Sheet. AEs occurring more than 30 days after last study treatment exposure date are not summarized. >>

### Table 14.3.1-6.7.1 Adverse events of interest incidence by specific group and preferred term during TFR phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the TFR phase

<< Programming note: Same shell as table 14.3.1-6.6.1 for TFR, use footnotes:</pre>

- Only adverse events from TFR phase are included in this table.
- Specific groups are alphabetically presented; preferred terms are sorted within each group in descending frequency of 'All grades' column. Percentage based on the number of patients included in the analysis population (N).
- Treatment Arm 1/Arm 2: 24/36 months, Re-treatment max Arm 1/Arm 2: 36/24 months.
- A patient with multiple occurrences of an AE is counted only once in the AE category. A patient with multiple AE within a primary system organ class is counted only once in the total row. AE of special interest CVEs (IHD), CVEs (PAOD), CVEs (ICD) and CVEs (others) are based on grouped MedDRA terms as described in the Case Retrieval Sheet. >>

### Table 14.3.1-6.7.2 Adverse events of interest occurrence by specific group and preferred term during TFR phase – overall and maximum grade 3/4 – Subset of Full Analysis Set entering the TFR phase

<< Programming note: Same shell as table 14.3.1-6.7.1 but without percentages use footnotes:</pre>

- Only adverse events from TFR phase are included in this table.
- Specific groups are alphabetically presented; preferred terms are sorted within each group in descending frequency of 'All grades' column.
- Treatment Arm 1/Arm 2: 24/36 months, Re-treatment max Arm 1/Arm 2: 36/24 months.
- AE of special interest CVEs (IHD), CVEs (PAOD), CVEs (ICD) and CVEs (others) are based on grouped MedDRA terms as described in the Case Retrieval Sheet.

# Table 14.3.1-7.1.1 Treatment Emergent adverse events of interest incidence, regardless of study drug relationship, by specific group and preferred term and by cardiovascular risk factors during Prerandomization Induction/consolidation phase – by treatment arm, overall and maximum grade 3/4 – Full Analysis Set

Very high or high risk / Moderate or low risk

| | Arm<br>N=x | | | m 2<br>xxx | | mized<br>xxx | | domized<br>xxx | | tal<br>xxx |
|---|---|---|---|---|---|---|---|---|---|---|
| Specific group<br>Preferred term | All grades<br>n (%) | Grade<br>3/4<br>n (%) | All<br>grades<br>n (%) | Grade<br>3/4<br>n (%) | All<br>grades<br>n (%) | Grade<br>3/4<br>n (%) | All<br>grades<br>n (%) | Grade<br>3/4<br>n (%) | All<br>grades<br>n (%) | Grade<br>3/4<br>n (%) |
| All AESI | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Group 1 | | | | | | | | | | |
| PT1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| • • • | | | | | | | | | | |
| Group 2 | | | | | | | | | | |
| PT1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

<sup>-</sup> Only TEAEs from pre-rand. ind./cons. phase are included in this table. Specific groups are presented alphabetically;

<sup>-</sup> PTs are sorted within each group in descending frequency of 'All grades' column.

<sup>-</sup> Percentage based on the population number (N). Treatment Arm 1/Arm 2: 24/36 months, Re-treatment max Arm 1/Arm 2: 36/24 months.

A patient with multiple occurrences of an AE is counted only once in the AE category.

<sup>-</sup> A patient with multiple AEs within a group is counted only once in the total row. AE of special interest CVEs (IHD), CVEs (PAOD), CVEs (ICD) and CVEs (others) are based on grouped MedDRA terms as described in the Case Retrieval Sheet.

<sup>-</sup> CV risk factors are defined as described in EU Guidelines on cardiovascular disease prevention in clin. Practice (version 2012). European Heart Journal (2012) 33, 1635-1701. AEs occurring more than 30 days after last study treatment exposure date are not summarized.

# Table 14.3.1-7.1.2 Treatment Emergent adverse events of interest occurrence, regardless of study drug relationship, by specific group and preferred term and by cardiovascular risk factors during Prerandomization Induction/consolidation phase – by treatment arm, overall and maximum grade 3/4 – Full Analysis Set

<< Programming note: Same shell as table 14.3.1-7.1.1 but without percentages use footnotes:</pre>

- Only TEAEs from pre-rand. ind./cons. phase are included in this table. Specific groups are presented alphabetically;
- PTs are sorted within each group in descending frequency of 'All grades' column.
- Treatment Arm 1/Arm 2: 24/36 months, Re-treatment max Arm 1/Arm 2:
- 36/24 months. AE of special interest CVEs (IHD), CVEs (PAOD), CVEs (ICD) and CVEs (others) are based on grouped MedDRA terms as described in the Case Retrieval Sheet.
- CV risk factors are defined as described in EU Guidelines on cardiovascular disease prevention in clinical practice (version 2012). European Heart Journal (2012) 33, 1635-1701. AEs occurring more than 30 days after last study treatment exposure date are not summarized.

# Table 14.3.1-7.2.1 Treatment-emergent adverse events of interest incidence, regardless of study drug relationship, during post-randomization consolidation phase (ARM 2), by specific group and preferred term, and by cardiovascular risk factor— overall and maximum grade 3 or 4 — Subset of Full Analysis Set randomized to Arm 2

7 mm 2

Subgroup: Cardiovascular risk factor at baseline: Very high/High risk (Note for programming: to be repeated on Moderate/Low risk)

Specific group

Preferred term

| Preferred term | N=xx | |
|---|---|---|
| | All grades<br>n (%) | Grade 3/4<br>n (%) |
| All AESI | xx (xx.x) | xx (xx.x) |
| Group 1<br>PT 1 | xx (xx.x) | xx (xx.x) |
| PT 2<br>ect | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) |
| Group 2 | | |
| PT 1 | xx (xx.x) | xx (xx.x) |
| PT 2 | xx (xx.x) | xx (xx.x) |
| ect | xx (xx.x) | xx (xx.x) |
| ect | | |

<sup>-</sup> Only TEAEs from post-rand. cons. phase are included in this table. Specific groups are presented alphabetically;
- PTs are sorted within each group in descending frequency of 'All grades' column. Percentage based on the population number (N). Treatment post-randomization Arm 2: 12 months, Re-treatment max Arm 2: 24 months. A patient with multiple occurrences of an AE is counted only once in the AE category. A patient with multiple AEs within a group is counted only once in the total row. AE of special interest CVEs (IHD), CVEs (PAOD), CVEs (ICD) and CVEs (others) are based on grouped MedDRA terms as described in the Case Retrieval Sheet. CV risk factors are defined as described in EU Guidelines on cardiovascular disease prevention in clin. practice (version 2012). European Heart Journal (2012) 33, 1635-1701. AEs occurring more than 30 days after last study treatment exposure date are not summarized.

<< Note for programming:

The "N" in header should correspond to the number of patient in the analysis set and in the selected cardiovascular risk factor subgroup.

When there is no patient in the analysis set and subgroup selected then do not display the subgroup.>>

# Table 14.3.1-7.2.2 Treatment-emergent adverse events of interest occurrence, regardless of study drug relationship, during post-randomization consolidation phase (ARM 2), by specific group and preferred term, and by cardiovascular risk factor – overall and maximum grade 3 or 4 – Subset of Full Analysis Set randomized to Arm 2

<< Programming note: Same shell as table 14.3.1-7.2.1 but without percentages use footnotes:</pre>

- Only TEAEs from post-rand. cons. phase are included in this table. Specific groups are presented alphabetically; PTs are sorted within each group in descending frequency of 'All grades' column.
- Treatment post-randomization Arm 2: 12 months, Re-treatment max Arm 2:
- 24 months. AE of special interest CVEs (IHD), CVEs (PAOD), CVEs (ICD) and CVEs (others) are based on grouped MedDRA terms as described in the Case Retrieval Sheet.
- CV risk factors are defined as described in EU Guidelines on cardiovascular disease prevention in clin. practice (version 2012). European Heart Journal (2012) 33, 1635-1701. AEs occurring more than 30 days after last study treatment exposure date are not summarized.

## Table 14.3.1-7.3.1 Treatment-emergent adverse events of interest incidence, regardless of study drug relationship, during re-treatment phase, by specific group and preferred term, and by cardiovascular risk factor – Subset of Full Analysis Set entering the re-treatment phase

Very high or high risk / Moderate or low risk

| | Arm | . 1 | Arm | 2 | Total | |
|---|---|---|---|---|---|---|
| | N=xxx | | | XX | N=xxx | |
| Specific group<br>Preferred term | All grades<br>n (%) | Grade<br>3/4<br>n (%) | All<br>grades<br>n (%) | Grade<br>3/4<br>n (%) | All<br>grades<br>n (%) | Grade<br>3/4<br>n (%) |
| All AESI | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Group 1 | | | | | | |
| PT1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ••• | | | | | | |
| Group 2 | | | | | | |
| PT1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

<sup>-</sup> Only TEAEs from re-treatment phase are included in this table. Specific groups are presented alphabetically;

<sup>-</sup> PTs are sorted within each group in descending frequency of 'All grades' column.

<sup>-</sup> Percentage based on the population number (N). Treatment Arm 1/Arm 2: 24/36 months, Re-treatment max Arm 1/Arm 2: 36/24 months. A patient with multiple occurrences of an AE is counted only once in the AE category. A patient with multiple AEs within a group is counted only once in the total row. AE of special interest CVEs (IHD), CVEs (PAOD), CVEs (ICD) and CVEs (others) are based on grouped MedDRA terms as described in the Case Retrieval Sheet. - CV risk factors are defined as described in EU Guidelines on cardiovascular disease prevention in clin. practice (version 2012). European Heart Journal (2012) 33, 1635-1701. AEs occurring more than 30 days after last study treatment exposure date are not summarized.

## Table 14.3.1-7.3.2 Treatment-emergent adverse events of interest occurrence, regardless of study drug relationship, during re-treatment phase, by specific group and preferred term, and by cardiovascular risk factor – Subset of Full Analysis Set entering the re-treatment phase

#### << Programming note: Same shell as table 14.3.1-7.3.1 but without percentages use footnotes:</pre>

- Only TEAEs from re-treatment phase are included in this table. Specific groups are presented alphabetically;
- PTs are sorted within each group in descending frequency of 'All grades' column.
- Treatment Arm 1/Arm 2: 24/36 months, Re-treatment max Arm 1/Arm 2: 36/24 months. AE of special interest CVEs (IHD), CVEs (PAOD), CVEs (ICD) and CVEs (others) are based on grouped MedDRA terms as described in the Case Retrieval Sheet.
- CV risk factors are defined as described in EU Guidelines on cardiovascular disease prevention in clin. practice (version 2012). European Heart Journal (2012) 33, 1635-1701. AEs occurring more than 30 days after last study treatment exposure date are not summarized.

## Table 14.3.1-7.4.1 Adverse events of interest incidence, regardless of study drug relationship, during TFR phase, by specific group and preferred term, and by cardiovascular risk factor – Subset of Full Analysis Set entering the TFR phase

<< Programming note: Same shell as table 14.3.1-7.3.1 for TFR, use footnotes:</pre>

- Only AEs from TFR phase are included in this table. Specific groups are presented alphabetically;
- PTs are sorted within each group in descending frequency of 'All grades' column.
- Percentage based on the population number (N). Treatment Arm 1/Arm 2: 24/36 months, Re-treatment max Arm 1/Arm 2: 36/24 months. A patient with multiple occurrences of an AE is counted only once in the AE category. A patient with multiple AEs within a group is counted only once in the total row. AE of special interest CVEs (IHD), CVEs (PAOD), CVEs (ICD) and CVEs (others) are based on grouped MedDRA terms as described in the Case Retrieval Sheet. CV risk factors are defined as described in EU on cardiovascular disease prevention in clin. practice (version 2012). European Heart Journal (2012) 33, 1635-1701. >>

## Table 14.3.1-7.4.2 Adverse events of interest occurrence, regardless of study drug relationship, during TFR phase, by specific group and preferred term, and by cardiovascular risk factor – Subset of Full Analysis Set entering the TFR phase

<< Programming note: Same shell as table 14.3.1-7.4.1 but without percentages, use footnotes:</pre>

- Only AEs from TFR phase are included in this table. Specific groups are presented alphabetically;
- PTs are sorted within each group in descending frequency of 'All grades' column.
- Treatment Arm 1/Arm 2: 24/36 months, Re-treatment max Arm 1/Arm 2:

36/24 months. AE of special interest CVEs (IHD), CVEs (PAOD), CVEs (ICD) and CVEs (others) are based on grouped MedDRA terms as described in the Case Retrieval Sheet. CV risk factors are defined as described in EU Guidelines on cardiovascular disease prevention in clin. practice (version 2012). European Heart Journal (2012) 33, 1635-1701.>>

- Table 14.3.1-7.5.1 Treatment-emergent adverse events of interest incidence, regardless of study drug relationship, during pre-randomization Induction/consolidation phase, by specific group and preferred term and by 4 cardiovascular risk factors overall and maximum grade 3/4 –Full Analysis Set
  - << Programming note: Same shell as table 14.3.1-7.1.1 but using: Very high risk, High risk, Moderate risk, Low risk>>
- Table 14.3.1-7.5.2 Treatment-emergent adverse events of interest occurence, regardless of study drug relationship, during pre-randomization Induction/consolidation phase, by specific group and preferred term and by 4 cardiovascular risk factors overall and maximum grade 3/4 –Full Analysis Set
  - << Programming note: Same shell as table 14.3.1-7.1.2 but using: Very high risk, High risk, Moderate risk, Low risk>>
- Table 14.3.1-7.6.1 Treatment-emergent adverse events of interest incidence, regardless of study drug relationship, during post-randomization consolidation phase (ARM 2), by specific group and preferred term, and by 4 categories of cardiovascular risk factors— overall and maximum grade 3 or 4 Subset of Full Analysis Set randomized to Arm 2
  - << Programming note: Same shell as table 14.3.1-7.2.1 but using: Very high risk, High risk, Moderate risk, Low risk>>
- Table 14.3.1-7.6.2 Treatment-emergent adverse events of interest occurrence, regardless of study drug relationship, during post-randomization consolidation phase (ARM 2), by specific group and preferred term, and by 4 categories of cardiovascular risk factors overall and maximum grade 3 or 4 Subset of Full Analysis Set randomized to Arm 2
  - << Programming note: Same shell as table 14.3.1-7.2.2 but using: Very high risk, High risk, Moderate risk, Low risk>>

- Table 14.3.1-7.7.1 Treatment-emergent adverse events of interest incidence, regardless of study drug relationship, during re-treatment phase, by specific group and preferred term, and by 4 categories of cardiovascular risk factors Subset of Full Analysis Set entering the re-treatment phase
  - << Programming note: Same shell as table 14.3.1-7.3.1 but using: Very high risk, High risk, Moderate risk, Low risk>>
- Table 14.3.1-7.7.2 Treatment-emergent adverse events of interest occurrence, regardless of study drug relationship, during re-treatment phase, by specific group and preferred term, and by 4 categories of cardiovascular risk factors— Subset of Full Analysis Set entering the re-treatment phase

<< Programming note: Same shell as table 14.3.1-7.3.2 but using: Very high risk, High risk, Moderate risk, Low risk>>

Table 14.3.1-7.8.1 Adverse events of interest incidence, regardless of study drug relationship, during TFR phase, by specific group and preferred term, and by 4 categories of cardiovascular risk factors – Subset of Full Analysis Set entering the TFR phase

<< Programming note: Same shell as table 14.3.1-7.4.1 but using: Very high risk, High risk, Moderate risk, Low risk>>

Table 14.3.1-7.8.2 Adverse events of interest occurrence, regardless of study drug relationship, during TFR phase, by specific group and preferred term, and by 4 categories of cardiovascular risk factors– Subset of Full Analysis Set entering the TFR phase

<< Programming note: Same shell as table 14.3.1-7.4.2 but using: Very high risk, High risk, Moderate risk, Low risk>>

### Table 14.3.1-9.1 On treatment deaths, by system organ class and preferred term during pre-randomization Induction/Consolidation phase - Safety Set

| Primary system organ class<br>Principal cause of death | Arm 1<br>N=xxx<br>n (%) | Arm 2<br>N=xxx<br>n (%) | Randomized<br>N=xxx<br>n (%) | Not Randomized<br>N=xxx<br>n (%) | Total<br>N=xxx<br>n (%) |
|---|---|---|---|---|---|
| Any Primary system organ class | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Primary system organ class 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred term 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred term 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| • • • | | • • • | • • • | • • • | |

<sup>-</sup> Primary system organ classes are alphabetically presented; preferred terms are sorted within primary system organ class in descending frequency.

<< Programming note: Include all deaths recorded on the AE CRF page>>

<sup>-</sup> Percentage based on the number of patients included in the analysis population (N).

<sup>-</sup> Treatment Arm 1/Arm 2: 24/36 months, Re-treatment max Arm 1/Arm 2: 36/24 months.

<sup>-</sup> Deaths up to 30 days after last study treatment exposure date are all included

<sup>-</sup> For patient # \_\_\_\_\_, date of death was imputed to " \_\_\_\_\_ ", from the original " \_\_\_\_ " for the purpose of this table only.

### Table 14.3.1-9.2 On treatment deaths, by system organ class and preferred term during post-randomization consolidation phase (ARM 2) – Subset of Safety Set randomized to Arm 2

| Primary system organ class<br>Principal cause of death | Arm 2<br>N=xxx<br>n (%) |
|---|---|
| Any Primary system organ class | xx (xx.x) |
| Primary system organ class 1 | xx (xx.x) |
| Preferred term 1 | xx (xx.x) |
| Preferred term 2 | xx (xx.x) |
| • • • | |

<sup>-</sup> Primary system organ classes are alphabetically presented; preferred terms are sorted within primary system organ class in descending frequency.

<<pre><<Pre>rogramming note: Include all deaths recorded on the AE CRF page>>

### Table 14.3.1-9.3 On treatment deaths, by system organ class and preferred term during re-treatment phase – Subset of Safety Set entering the re-treatment phase

<< Programming note: Same shell as table 14.3.1-9.1 presenting only Arm 1, Arm 2 and Total, use footnotes:>

Primary system organ classes are alphabetically presented; preferred terms are sorted within primary system organ class in descending frequency.

- Only deaths occurring during the treatment period (between the first day of study drug intake and up to 30 days after last study drug intake) are presented.
- Percentage based on the number of patients included in the analysis population (N).
- Treatment Arm 1/Arm 2: 24/36 months, Re-treatment max Arm 1/Arm 2: 36/24 months.

<sup>-</sup> Percentage based on the number of patients included in the analysis population (N).

<sup>-</sup> Treatment post-randomization Arm 2: 12 months, Re-treatment max Arm 2: 24 months.

<sup>-</sup> Deaths up to 30 days after last study treatment exposure date are all included

Table 14.3.1-10.1.1 Cardiac and vascular adverse events of interest, incidence, by treatment arm during the pre-randomization induction/consolidation phase - Full Analysis Set

| | Ar | m 1 | Ar | m 1 | Rand | lomized | Not Rar | ndomized | Тс | tal |
|---|---|---|---|---|---|---|---|---|---|---|
| | N= | XXX | N= | XXX | N: | =xxx | N= | XXX | N= | ××× |
| Cardiac and vascular | All<br>grades | Grade<br>3/4 | All<br>grades | Grade<br>3/4 | All<br>grades | Grade 3/4 | All<br>grades | Grade<br>3/4 | All<br>grades | Grade<br>3/4 |
| adverse events | n (%) | n (%) | n (%) | n (%) | n (%) | . , | n (%) | n (%) | n (%) | n (%) |
| Any cardiac event | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any serious cardiac event | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any cardiac event related to study treatment | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any cardiac event leading<br>to study drug<br>discontinuation | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any vascular event | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any serious vascular event | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any vascular event related to study treatment | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any vascular event<br>leading to study drug<br>discontinuation | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of cardiac events per patient | | | | | | | | | | |
| 0 time | XX | xx | xx | XX | XX | XX | XX | XX | XX | XX |
| 1 time | XX | XX | XX | XX | XX | XX | xx | XX | xx | xx |

|---|---|---|---|---|---|---|---|---|---|---|
| RAP Module 7.1 | | | 6- | May-2021 (14 | 1:35) | | | Protocol No CAMN107AIC0 | | |
| 2 times | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| 3 times | XX | xx | XX | XX | XX | XX | XX | XX | XX | xx |
| 4 or more times | XX | XX | XX | XX | XX | XX | XX | XX | XX | xx |
| Number of vascular event per patient | S | | | | | | | | | |
| 0 time | XX | xx | XX | xx | XX | XX | XX | XX | XX | xx |
| 1 time | XX | xx | XX | xx | XX | XX | XX | XX | XX | xx |
| 2 times | XX | XX | XX | XX | XX | XX | XX | XX | XX | xx |
| 3 times | XX | XX | XX | XX | XX | XX | XX | XX | xx | XX |
| 4 or more times | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |

<sup>-</sup> Only pre-randomization events occurring during induction/consolidation or within 30 days after the last study treatment exposure (pre-randomization consolidation period 12-24 months) date are displayed. Percentage based on the number of patients included in the analysis population (N).

<<pre><<Pre>rogramming note: Only adverse events of special interest are displayed, there are defined with case retrieval sheet where
compound are: CVES(IHD), CVEs (PAOD), CVEs (ICD) and CVEs (others) (AEVSG not empty in A\_AEV dataset and SOC= Cardiac
disorders or Vascular disorders). If date of start of AE \leq Day 365 then AE will be count in induction phase, else if date of
start of AE > Day 365 then it will be considered in consolidation phase. >>

<sup>-</sup> Treatment Arm 1/Arm 2: 24/36 months, Re-treatment max Arm 1/Arm 2: 36/24 months. A patient with multiple occurrences of an event is counted only once. Events of interest CVEs (IHD), CVEs (PAOD), CVEs (ICD) and CVEs (others) are based on grouped MedDRA terms from the Case Retrieval Sheet. Cardiac events correspond to events of interest with System Organ Class "Cardiac disorders" and vascular events correspond to events of interest with System Organ Class "Vascular disorders".

### Table 14.3.1-10.1.2 Cardiac and vascular adverse events of interest, occurrence, by treatment arm during the pre-randomization induction/consolidation phase - Full Analysis Set

<< Programming note: Same shell as table 14.3.1-10.1.1 but without percentages, use footnotes:

- Only pre-randomization events occurring during induction/consolidation or within 30 days after the last study treatment exposure (pre-randomization consolidation period 12-24 months) date are displayed.
- Treatment Arm 1/Arm 2: 24/36 months, Re-treatment max Arm 1/Arm 2: 36/24 months. Events of interest CVEs (IHD), CVEs (PAOD), CVEs (ICD) and CVEs (others) are based on grouped MedDRA terms from the Case Retrieval Sheet. Cardiac events correspond to events of interest with System Organ Class "Cardiac disorders" and vascular events correspond to events of interest with System Organ Class "Vascular disorders".

Table 14.3.1-10.2.1 Cardiac and vascular adverse events of interest incidence, during the post-randomization consolidation phase (ARM 2) - Subset of Full Analysis Set randomized to Arm 2

| | Ar | m 2 |
|---|---|---|
| | N= | XXX |
| Cardiac and vascular | All<br>grades | Grade<br>3/4 |
| adverse events | n (%) | n (%) |
| Any cardiac event | xx (xx.x) | xx (xx.x) |
| Any serious cardiac event | xx (xx.x) | xx (xx.x) |
| Any cardiac event related to study treatment | xx (xx.x) | xx (xx.x) |
| Any cardiac event leading to study drug discontinuation | xx (xx.x) | xx (xx.x) |
| Any vascular event | xx (xx.x) | xx (xx.x) |
| Any serious vascular event | xx (xx.x) | xx (xx.x) |
| Any vascular event related to study treatment | xx (xx.x) | xx (xx.x) |
| Any vascular event leading to study drug discontinuation | xx (xx.x) | xx (xx.x) |
| Number of cardiac events per patient | | |
| 0 time | XX | xx |
| 1 time | XX | xx |
| 2 times | XX | xx |
| 3 times | XX | xx |
| 4 or more times | XX | XX |
| Number of vascular events per patient | | |
| 0 time | XX | XX |

| Novartis<br>RAP Module 7.1 | Confidential<br>6-May-2021 (14:35) | Page 381<br>Protocol No CAMN107AIC0 |
|---|---|---|
| 1 time | xx xx | |
| 2 times | xx xx | |
| 3 times | xx xx | |
| 4 or more times | XX XX | |

- Only events occurring during post-randomization or within 30 days after the last study treatment exposure (post-randomization consolidation period 12 months) date are displayed. Percentage based on the number of patients included in the analysis population (N).
- Treatment post-randomization Arm 2: 12 months. A patient with multiple occurrences of an event is counted only once. Events of interest CVEs (IHD), CVEs (PAOD), CVEs (ICD) and CVEs (others) are based on grouped MedDRA terms from the Case Retrieval Sheet. Cardiac events correspond to events of interest with System Organ Class "Cardiac disorders" and vascular events correspond to events of interest with System Organ Class "Vascular disorders".

### Table 14.3.1-10.2.2 Cardiac and vascular adverse events of interest occurrence, during the post-randomization consolidation phase (ARM 2) - Subset of Full Analysis Set randomized to Arm 2

<< Programming note: Same shell as table 14.3.1-10.2.1 but without percentages, use footnotes:

- Only events occurring during post-randomization or within 30 days after the last study treatment exposure (post-randomization consolidation period 12 months) date are displayed.
- Treatment post-randomization Arm 2: 12 months. Events of interest CVEs (IHD), CVEs (PAOD), CVEs (ICD) and CVEs (others) are based on grouped MedDRA terms from the Case Retrieval Sheet. Cardiac events correspond to events of interest with System Organ Class "Cardiac disorders" and vascular events correspond to events of interest with System Organ Class "Vascular disorders".

### Table 14.3.1-10.3.1 Cardiac and vascular adverse events of interest, incidence, by treatment arm during the retreatment phase – Subset of Full Analysis Set entered re-treatment phase

<< Programming note: Same shell as table 14.3.1-10.1.1 but for re-treatment, use footnotes:

- Only events occurring during re-treatment phase or within 30 days after the last study treatment exposure (re-treatment period 24-36 months) date are displayed. Percentage based on the number of patients included in the analysis population (N).
- Treatment Arm 1/Arm 2: 24/36 months, Re-treatment max Arm 1/Arm 2: 36/24 months. A patient with multiple occurrences of an event is counted only once. Events of interest CVEs (IHD), CVEs (PAOD), CVEs (ICD) and CVEs (others) are based on grouped MedDRA terms from the Case Retrieval Sheet. Cardiac events correspond to events of interest with System Organ Class "Cardiac disorders" and vascular events correspond to events of interest with System Organ Class "Vascular disorders".

### Table 14.3.1-10.3.2 Cardiac and vascular adverse events of interest, occurrence, by treatment arm during the re-treatment phase - Subset of Full Analysis Set entered re-treatment phase

- << Programming note: Same shell as table 14.3.1-10.3.1 but without percentages, using footnotes:</pre>
- Only events occurring during re-treatment phase or within 30 days after the last study treatment exposure (re-treatment period 24-36 months) date are displayed.
- Treatment Arm 1/Arm 2: 24/36 months, Re-treatment max Arm 1/Arm 2: 36/24 months. Events of interest CVEs (IHD), CVEs (PAOD), CVEs (ICD) and CVEs (others) are based on grouped MedDRA terms from the Case Retrieval Sheet. Cardiac events correspond to events of interest with System Organ Class "Cardiac disorders" and vascular events correspond to events of interest with System Organ Class "Vascular disorders".
### Table 14.3.1-10.4.1 Cardiac and vascular adverse events of interest, incidence, by treatment arm during the TFR phase – Subset of Full Analysis Set entered TFR phase

<< Programming note: Same shell as table 14.3.1-10.1.1 but for TFR use footnotes:</pre>

- Only events occurring during TFR phase (TFR period 24-36 months) date are displayed.
- Percentage based on the number of patients included in the analysis population (N).
- Treatment Arm 1/Arm 2: 24/36 months, Re-treatment max Arm 1/Arm 2: 36/24 months.
- A patient with multiple occurrences of an event is counted only once.
- Events of interest CVEs (IHD), CVEs (PAOD), CVEs (ICD) and CVEs (others) are based on grouped MedDRA terms from the Case Retrieval Sheet. Cardiac events correspond to events of interest with System Organ Class "Cardiac disorders" and vascular events correspond to events of interest with System Organ Class "Vascular disorders".>>

### Table 14.3.1-10.4.2 Cardiac and vascular adverse events of interest, occurrence, by treatment arm during the TFR phase - Subset of Full Analysis Set entered TFR phase

 $<\!<\!Programming\ note:\ Same\ shell\ as\ table\ 14.3.1-10.4.1\ but\ without\ percentages\ use\ footnotes:$ 

- Only events occurring during TFR phase (TFR period 24-36 months) date are displayed.
- Treatment Arm 1/Arm 2: 24/36 months, Re-treatment max Arm 1/Arm 2: 36/24 months.
- Events of interest CVEs (IHD), CVEs (PAOD), CVEs (ICD) and CVEs (others) are based on grouped MedDRA terms from the Case Retrieval Sheet. Cardiac events correspond to events of interest with System Organ Class "Cardiac disorders" and vascular events correspond to events of interest with System Organ Class "Vascular disorders".>>

Table 14.3.1-10.5 Relationship between cardiac and vascular adverse events of interest with total cholesterol values - Full Analysis Set

| | Total Cholesterol Values | | | |
|---|---|---|---|---|
| Adverse events | <= 5.2 mmol/L | >5.2 and $<=6.2$ mmol/L | > 6.2 mmol/L | Missing |
| Cardiac events | | | | |
| Yes | XX | XX | XX | XX |
| No | XX | xx | XX | XX |
| Vascular events | | | | |
| Yes | XX | XX | XX | XX |
| No | XX | XX | XX | XX |

<sup>-</sup> All events are considered, even if occurred on same patient. All AEs occurring during the study or within 30 days after the last study treatment exposure date are displayed. For patients with event, the last laboratory available assessment before or at date of start of the event is considered. When the date of the AE is missing, the first laboratory assessment after the start of the study med. is considered. Patients without event are counted only once, presented under the highest total cholesterol value. Events of interest CVEs (IHD), CVEs (PAOD), CVEs (ICD) and CVEs (others) are based on grouped MedDRA terms from the Case Retrieval Sheet. Cardiac events correspond to events of interest with SOC "Cardiac disorders" and vascular events correspond to events of interest with SOC "Vascular disorders".

<<Pre><<Pre>rogramming note: Only adverse events of special interest are displayed, there are defined with case retrieval sheet where
compound are: CVES(IHD), CVEs (PAOD), CVEs (ICD) and CVEs (others) (AEVSG not empty in A\_AEV dataset and SOC= Cardiac
disorders or Vascular disorders).

Patient with no event of interest should be counted in category NO of highest value post-baseline or in category Missing otherwise.>>

Table 14.3.1-10.6 Relationship between cardiac and vascular adverse events of interest with glycemic values - Full Analysis Set

| | Fasting Glucose Values | | |
|-----------------|------------------------|--------------|---------|
| Adverse events | ≤6.9 mmol/L | > 6.9 mmol/L | Missing |
| Cardiac events | | | |
| Yes | XX | xx | XX |
| No | XX | XX | XX |
| Vascular events | | | |
| Yes | xx | XX | XX |
| No | XX | XX | XX |

- All events are considered, even if occurred on same patient. All AEs during the study or within 30 days after the last study treatment exposure date are displayed. For patients with event, the last laboratory available assessment before or at date of start of the first event is considered. When the date of the AE is missing, the first laboratory assessment after the start of the study med. is considered. Patients without event are counted only once, presented under the highest fasting glucose value. Events of interest CVEs (IHD), CVEs (PAOD), CVEs (ICD) and CVEs (others) are based on grouped MedDRA terms from the Case Retrieval Sheet. Cardiac events correspond to events of interest with SOC "Cardiac disorders" and vascular events correspond to events of interest with SOC "Vascular disorders".

<<pre><<Pre>rogramming note: Only adverse events of special interest are displayed, there are defined with case retrieval sheet where
compound are: CVES(IHD), CVEs (PAOD), CVEs (ICD) and CVEs (others) (AEVSG not empty in A\_AEV dataset and SOC= Cardiac
disorders or Vascular disorders).>>

Table 14.3.1-11.1.1 Kaplan-Meier estimate of time-to-first CVEs during the pre-randomization induction/consolidation phase – Full analysis set

| KM estimates | Arm 1<br>N=xx | Arm 2<br>N=xx | Randomized<br>N=xx | Not<br>Randomized<br>N=xx | Total<br>N=xx |
|---|---|---|---|---|---|
| Number of patients - n (%) | | | | | |
| with events | xxx (xx.x) | xxx (xx.x) | | | xxx (xx.x) |
| with censorings | xxx (xx.x) | xxx (xx.x) | | | xxx (xx.x) |
| Time to event (months) | | | | | |
| 25th percentile (95% CI) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) | | | xx.x (xx.x, xx.x) |
| Median (95% CI) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) | • • • | • • • | xx.x (xx.x, xx.x) |
| 75 <sup>th</sup> percentile (95% CI) | xx.x (xx.x, xx.x) | xx.x ( $xx.x$ , $xx.x$ ) | • • • | | xx.x ( $xx.x$ , $xx.x$ ) |
| Percentage of patients | | | | | |
| without event - | | | | | |
| Estimate (95% CI) | | | | | |
| 6 months | xx.x $(xx.x)$ $(xx.x, xx.x)$ | xx.x(xx.x) $(xx.x, xx.x)$ | | | xx.x(xx.x) $(xx.x, xx.x)$ |
| 12 months | xx.x (xx.x) xx.x, xx.x) | xx.x(xx.x) (xx.x, xx.x) | | | xx.x(xx.x) (xx.x, xx.x) |
| 18 months | xx.x (xx.x) (xx.x, xx.x) | xx.x(xx.x) (xx.x, xx.x) | | | xx.x(xx.x) (xx.x, xx.x) |
| 24 months | xx.x ( $xx.x$ ) ( $xx.x$ , $xx.x$ ) | xx.x(xx.x) (xx.x, xx.x) | | | xx.x(xx.x) $(xx.x, xx.x)$ |

<sup>-</sup> NE: Not Estimable.

<sup>-</sup> Event = first occurrence of CVE during the pre-randomization induction/consolidation phase.

<sup>-</sup> Censoring rule = patients who did not meet the event are censored to the minimum date between the last contact date, the end of induction/consolidation phase, the randomization date the date of death.

<sup>-</sup> n is the number of patients at risk at the timepoint (i.e. without event and still ongoing)

<sup>-</sup> The percentage of patients without event and the respective 95% C.I. are estimated from Kaplan Meier.

<sup>-</sup> Presenting CVEs occurred within Pre-Randomization Ind/Cons phase only, excluding additional +30 days period used in TEAE outputs.

```
proc lifetest data=data outsurv=surv stderr method=km atrisk;
  time VART*evt(0);
  strata TRT;
    ods output
    Quartiles =Quartile
    ProductLimitEstimates=lifetable
    censoredsummary=Censum(keep=TRT stratum failed total censored);
*Frame for all time points (please use maximum time as required. As an example here I am using 1-50);
data frame;
  do TRT= 1 to 2;
   do VART= 1 to 50 by 1;
      output;
   end:
  end;
run;
proc sort data=frame ; by TRT VART; run;
proc sort data=surv ; by TRT VART; run;
data surv1;
  merge surv(in=a) frame(in=b);
  if a or b;
  by TRT VART;
********Using LOCF to impute all records with valid results ******;
data surv2;
   set surv1;
   retain psurv up low;
  by TRT;
   if first.TRT then psurv=.;
   if survival ne . then psurv=survival;
   if first.TRT then up=.;
   if sdf ucl ne . then up=sdf ucl;
   if first.TRT then low=.;
   if sdf lcl ne . then low=sdf lcl;
 run:
*Keep only 1 row per time point per treatment arm. Find specific timepoint;
```

Novartis Confidential Page 388 RAP Module 7.1 6-May-2021 (14:35) Protocol No CAMN107AIC0

proc sort data=surv2 out=surv3 nodupkey; by TRT VART; run;
\*Quartile and Censum contain the information for the first two parts of the table;

## Table 14.3.1-11.1.2 Kaplan-Meier estimate of time-to-first CVEs during the post-randomization consolidation phase (ARM 2)— Subset of Full Analysis Set patients randomized on Arm 2

| KM estimates | Arm2<br>N=xx |
|---|---|
| Number of patients - n (%) with events | xxx (xx.x) |
| with censorings | xxx (xx.x) |
| Time to event (months) | |
| 25th percentile (95% CI) | xx.x (xx.x, xx.x) |
| Median (95% CI) | xx.x (xx.x, xx.x) |
| 75 <sup>th</sup> percentile (95% CI) | xx.x ( $xx.x$ , $xx.x$ ) |
| Percentage of patients without event - Estimate n(%) (95% CI) | |
| 6 months | xx.x (xx.x) (xx.x, xx.x) |
| 12 months | xx.x(xx.x) $(xx.x, xx.x)$ |

<sup>-</sup> NE: Not Estimable.

<sup>-</sup> Event = first occurrence of CVE during the post-randomization induction/consolidation phase.

<sup>-</sup> Censoring rule = patients who did not meet the event are censored to the minimum date between the last contact date, the end of induction/consolidation phase and the date of death.

<sup>-</sup> n is the number of patients at risk at the timepoint (i.e. without event and still ongoing)

<sup>-</sup> The percentage of patients without event and the respective 95% C.I. are estimated from Kaplan Meier.

<sup>-</sup> Patients randomized to Arm 2 have 12 months of treatment post-randomization and a maximum of 24 months of re-treatment.

<sup>-</sup> Presenting CVEs occurred within Post-Randomization consolidation phase only, excluding additional +30 days period used in TEAE outputs.

Table 14.3.1-11.2 Kaplan-Meier estimate of time-to-first CVEs during the re-treatment phase – Subset of Full Analysis Set entering the re-treatment phase

| KM estimates | Arm 1<br>N=xx | Arm 2<br>N=xx | Total<br>N=xx |
|---|---|---|---|
| Number of patients - n (%) | | | |
| with events | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| with censorings | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Time to event (months) | | | |
| 25th percentile (95% CI) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| Median (95% CI) | xx.x ( $xx.x$ , $xx.x$ ) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| 75 <sup>th</sup> percentile (95% CI) | xx.x ( $xx.x$ , $xx.x$ ) | xx.x (xx.x, xx.x) | xx.x ( $xx.x$ , $xx.x$ ) |
| Percentage of patients without event - | | | |
| Estimate n(%) (95% CI) | | | |
| 6 months | xx.x $(xx.x)$ $(xx.x, xx.x)$ | xx.x ( $xx.x$ ) ( $xx.x$ , $xx.x$ ) | xx.x (xx.x) (xx.x, xx.x) |
| 12 months | xx.x ( $xx.x$ ) ( $xx.x$ , $xx.x$ ) | xx.x ( $xx.x$ ) ( $xx.x$ , $xx.x$ ) | xx.x (xx.x) (xx.x, xx.x) |
| 24 months | xx.x ( $xx.x$ ) ( $xx.x$ , $xx.x$ ) | xx.x $(xx.x)$ $(xx.x, xx.x)$ | xx.x (xx.x) (xx.x, xx.x) |
| 30 months | xx.x $(xx.x)$ $(xx.x, xx.x)$ | | xx.x $(xx.x)$ $(xx.x, xx.x)$ |
| 36 months | xx.x $(xx.x)$ $(xx.x, xx.x)$ | | xx.x (xx.x) (xx.x, xx.x) |

- NE: Not Estimable.
- Event = first occurrence of CVE during the re-treatment phase.
- Censoring rule = patients who did not meet the event are censored to the minimum date between the last contact date, the end of re-treatment phase and the date of death.
- n is the number of patients at risk at the timepoint (i.e. without event and still ongoing)
- The percentage of patients without event and the respective 95% C.I. are estimated from Kaplan Meier.
- Patients randomized to Arm 1 have 24 months of treatment and a maximum of 36 months of re-treatment.
  - Patients randomized to Arm 2 have 36 months of treatment and a maximum of 24 months of re-treatment.
- Presenting CVEs occurred within Re-treatment phase only, excluding additional +30 days period used in TEAE outputs.

#### << Programming note: Time to start date is the first day of re-treatment phase.>>

Table 14.3.1-12.1 Medical history by system organ class and preferred term- Full Analysis Set

| System organ class<br>Preferred term | Arm 1<br>N=xxx<br>n(%) | Arm 2<br>N=xxx<br>n(%) | Randomized<br>N=xxx<br>n(%) | Not Randomized<br>N=xxx<br>n(%) | Total<br>N=xxx<br>n(%) |
|---|---|---|---|---|---|
| SOC1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT1<br>PT2 | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br> | xx (xx.x)<br>xx (xx.x) |
| SOC2 | xx (xx.x)<br> | xx (xx.x)<br> | xx (xx.x)<br> | xx (xx.x)<br> | xx (xx.x)<br> |

<sup>-</sup> Primary system organ classes are presented alphabetically; preferred terms are sorted within Primary system organ class by descending frequency.

Table 14.3.1-13.1 Prior exposure to imatinib before screening, MMR, age, and Sokal by LSC detection category - LSC sub-study Full Analysis Set

Baseline#

| | | LSC | detected | LSC not detected | |
|---|---|---|---|---|---|
| | | | n (응) | n | (%) |
| | | Not<br>Randomized<br>N=XX | Randomized<br>(Arm 1 and Arm 2)<br>N=XX | Not<br>Randomized<br>N=XX | Randomized<br>(Arm 1 and Arm 2)<br>N=XX |
| Prior Imatinib exposure | <5 years | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | >= 5 years | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| MMR | Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Age | <65 years | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | >= 65 years | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Sokal score | Low risk | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Intermediate risk | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | High risk | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

<sup>-</sup> LSC detected defined as Ph+ CD34/38+, or CD34/CD38-, or Immunophenotypically aberrant CD34+, or Immunophenotypically aberrant CD34-, for HIS, or PCR, or both.

Programming Note: Separate denominator for each column. Percentages sum up to 100% for each column/variable.

<sup>#</sup> Baseline value, latest available valid evaluation between Screening and Rescreening.

Table 14.3.1-13.2.1 Percentage from total CD34+ cells, CD34+/CD38+ cells - Subgroup of LSC sub-study Full Analysis Set, LSC detected

| | LSC<br>cells | Arm 1<br>(N=xx) | Arm 2<br>(N=xx) | Randomized (Arm 1 and Arm 2) (N=xx) | Not Randomized (N=xx) | Total (Randomized and Not Randomized) (N=xx) |
|---|---|---|---|---|---|---|
| Baseline# | n | xxx | xxx | xxx | xxx | xxx |
| 200011110 | Mean | xx.x | XX.X | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | X.XX | X.XX | X.XX |
| | 25 <sup>th</sup> percentile | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Median | xx.x | XX.X | XX.X | XX.X | XX.X |
| | 75 <sup>th</sup> percentile | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | xx.x, xx.x | xx.x, xx.x | XX.X, XX.X | xx.x, xx.x | xx.x, xx.x |
| Month 24 | n | XXX | XXX | XXX | xxx | xxx |
| | Min, Max | XX.X, XX.X | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Change from Baseline<br>to Month 24 | n | xxx | xxx | xxx | xxx | xxx |
| | Min, Max | XX.X, XX.X | XX.X, XX.X | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Month 36* | n | xxx | XXX | xxx | xxx | XXX |
| | | | • • • | | • • • | • • • |
| | Min, Max | xx.x, xx.x | XX.X, XX.X | xx.x, xx.x | XX.X, XX.X | XX.X, XX.X |
| Change from Baseline<br>to Month 36* | n | | XXX | | | xxx |
| | • • • | | • • • | | | • • • |
| | Min, Max | | xx.x, xx.x | | | xx.x, xx.x |

|----------------|--------------------|-------------------------|
| RAP Module 7.1 | 6-May-2021 (14:35) | Protocol No CAMN107AIC0 |

| EOP TFR | n | xxx | xxx | xxx | xxx |
|---|---|---|---|---|---|
| | Min, Max | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Change from Baseline<br>to EoP TFR | n | xxx | xxx | xxx | xxx |
| | Min, Max | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |

<sup>-</sup> LSC detected defined as Ph+ CD34/38+, or CD34/CD38-, or Immunophenotypically aberrant CD34+, or Immunophenotypically aberrant CD34-, for HIS, or PCR, or both.

# Table 14.3.1-13.2.2 Percentage from total CD34+ cells, CD34+/CD38- cells - Subgroup of LSC sub-study Full Analysis Set, LSC detected

<< Programming note: Same shell as Table 14.3.1-13.2.1 >>

# Table 14.3.1-13.2.3 Percentage from total CD34+ cells, Immunophenotypically aberrant CD34+ cells - Subgroup of LSC sub-study Full Analysis Set, LSC detected

<< Programming note: Same shell as Table 14.3.1-13.2.1 >>

<sup>#</sup> Baseline value, latest available valid evaluation between Screening and Rescreening.

<sup>\*</sup> For subjects randomized to Arm 2.

Table 14.3.1-13.2.4 Percentage from total CD34+ cells, Immunophenotypically aberrant CD34 negative cells - Subgroup of LSC sub-study Full Analysis Set, LSC detected

<< Programming note: Same shell as Table 14.3.1-13.2.1>>

Table 14.3.1-13.3.1 Percentage of Ph+ cells, CD34+/CD38- cells - Subgroup of LSC sub-study Full Analysis Set, LSC detected

<< Programming note: Same shell as Table 14.3.1-13.2.1>>

Table 14.3.1-13.3.2 Percentage of Ph+ cells, CD34+/CD38- cells - Subgroup of LSC sub-study Full Analysis Set, LSC detected

<< Programming note: Same shell as Table 14.3.1-13.2.1>>

Table 14.3.1-13.3.3 Percentage of Ph+ cells, Immunophenotypically aberrant CD34+ cells - Subgroup of LSC sub-study Full Analysis Set, LSC detected

<< Programming note: Same shell as Table 14.3.1-13.2.1>>

Table 14.3.1-13.3.4 Percentage of Ph+ cells, Immunophenotypically aberrant CD34 negative cells - Subgroup of LSC sub-study Full Analysis Set, LSC detected

<< Programming note: Same shell as Table 14.3.1-13.2.1>>

Table 14.3.1-13.4 Total Percentage of CD34+ cells- Subgroup of LSC sub-study Full Analysis Set, LSC detected

<< Programming note: Same shell as Table 14.3.1-13.2.1>>

Table 14.3.1-13.5 LSC detection - LSC sub-study Full Analysis Set

| | LSC<br>detected | Arm 1<br>(N=xx)<br>n(%) | Arm 2<br>(N=xx)<br>n(%) | Randomized (Arm 1 and Arm 2) (N=xx) n(%) | Not Randomized (N=xx) n(%) | Total (Randomized ar Not Randomized (N=xx) n(%) |
|---|---|---|---|---|---|---|
| Baseline# | Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Missing | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Month 24 | Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Missing | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Month 36* | Yes | | xx (xx.x) | | xx (xx.x) | xx (xx.x) |
| | No | | xx (xx.x) | | xx (xx.x) | xx (xx.x) |
| | Missing | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| EoP TFR | Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Missing | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

<sup>-</sup> LSC detected defined as Ph+ CD34/38+, or CD34/CD38-, or Immunophenotypically aberrant CD34+, or Immunophenotypically aberrant CD34-, for HIS, or PCR, or both.

<sup>#</sup> Baseline value, latest available valid evaluation between Screening and Rescreening.

<sup>\*</sup>For subjects randomized to Arm 2.

### Section 14.3.2 – Listings of deaths, other serious and significant adverse events

### Listing 14.3.2-1.1 Listing of deaths – Full Analysis Set

| Country/<br>Center/<br>Patient/<br>Arm | Age/<br>Sex/<br>Race | Date of<br>last dose | Study<br>day of<br>last<br>dose | Date of death (phase) | Study day<br>of death | Number days<br>since last<br>dose | Principal cause of<br>death reported/<br>Preferred term |
|---|---|---|---|---|---|---|---|
| XXX/0XXX/0XXXX/X | XX/X/XX | DDMMMYYYY | XX | DDMMMYYYY<br>(IND/CONS1/CONS2/TFR/<br>RE-TRT) | XX | xx | XXXXXXXXX/XXXXXX |
| XXX/0XXX/0XXXX/X@ | XX/X/XX | DDMMMYYYY | XX | DDMMMYYYY<br>(IND/CONS1/CONS2/TFR/<br>RE-TRT) | xx # | xx * | XXXXXXXXX/XXXXXX |

<sup>-</sup> Arm: 1: Arm 1; 2: Arm 2; 3: Not Randomized. - Phase: IND = ind. phase (0-12 m), CONS1 = pre-rand. Cons. Phase (12-24 m), CONS2 = post-rand. Cons phase (ARM 2)(24-36 m), TFR=Treat. free remission phase and RE-TRT=re-treat. phase. The phase displayed indicates in which end of phase page the death has been recorded as the primary reason to discontinue the study. If missing then death has been recorded in survival follow-up CRF pages.

- Study day relative to the first day of treatment (day 1).
- \* Event occurred more than 30 days after last study treatment exposure date.
- # Death occurring outside the treatment emergent period.
- @ For patient # death occurred during Survival follow-up.
- Number of days since last dose = day of death day of last dose + 1.

### Listing 14.3.2-1.2 Listing of deaths SDV sensitivity – Full Analysis Set

<< Programming note: Same shell as Listing 14.3.2-1.1, for SDV sensitivity analysis>>
Add footnote:

- SDV sensitivity: Excluding patient visits involved in SDV issues during final data review due to COVID-19

#### Listing 14.3.2-2.1 Listing of adverse events of special interest – Full Analysis Set

| Country/<br>Center/<br>Patient/<br>Arm | Age/<br>Sex/<br>Race | Adverse Event Verbatim/ Abbreviated System organ class/ Preferred term | Start date<br>/day | End date<br>/day | Dur<br>(days) | Phase | Grade/Relation/<br>Action taken |
|---|---|---|---|---|---|---|---|
| | /1 | Verbatim/Ab SOCxxxxxx / PTxxxxxxxxxxx | 16JUL2005/-2^ | 27JUL2005/13 | 12 | IC | G1/NS/A0 |
| | | Verbatim/Ab SOCxxxxxx /<br>PTxxxxxxxxxxx | 18JUL2005/4 | 27JUL2005/13 | 10 | TFR | G1/S/A3,5 |
| | /2 | Verbatim/Ab SOCxxxxxx /<br>PTxxxxxxxxxxxx | 16JUL2005/-1* | 27JUL2005/13 | 12 | RE-TRT | G1/NS/A0 |

- Arm: 1: Arm 1; 2: Arm 2; 3: Not Randomized.
- Phase: IC=Induction/Consolidation phase, TFR=TFR phase and RE-TRT=Re-treatment phase
- Relationship to study drug: NS=Not suspected, S=Suspected.
- Action taken: A0=No action taken, A1=Study drug dosage adjusted/temporarily interrupted, A2=Study drug permanently discontinued due to this AE, A3=Concomitant medication taken, A4=Non-drug therapy given, A5=Hospitalization/Prolonged hospitalization.
- Day is relative to the first day of treatment (day 1).
- \* Event occurred more than 30 days after the last study treatment exposure date. ^ Event occurred between patient's informed consent date and the day before first dose of study medication.

### Listing 14.3.2-2.2 Listing of adverse events leading to study drug discontinuation – Full Analysis Set

<< Programming note: Same shell as listing 14.3.2-2.1 on adverse events leading to study drug discontinuation >>

- Arm: 1: Arm 1; 2: Arm 2; 3: Not Randomized. Phase: IC=Induction/Consolidation phase, TFR=TFR phase and RE-TRT=Re-treatment phase. Relationship to study drug: NS=Not suspected, S=Suspected.
- Action taken: A0=No action taken, A1=Study drug dosage adjusted/temporarily interrupted, A2=Study drug permanently discontinued due to this AE, A3=Concomitant medication taken, A4=Non-drug therapy given, A5=Hospitalization/Prolonged hospitalization. Day is relative to the first day of treatment (day 1).
- \* Event occurred more than 30 days after the last study treatment exposure date. ^ Event occurred between patient's informed consent date and the day before first dose of study medication.
- Patient # reported as disc. Ind/Cons phase due to AE "Blast Crisis"- G2, should have been reported as disc. Ind/Cons phase due to Disease Progression, progression to Blast Crisis, as per Prot.

#### Add following footnote at the end of last page:

- For patient # due to reconciliation discrepancies, safety database reported AE term "Endometriosis" as a SAE, while in clinical database this AE was not recorded as an SAE.

## Listing 14.3.2-2.3 Listing of adverse events leading to study drug discontinuation during re-treatment phase – Subset of Full Analysis Set entering the re-treatment period

<< Programming note: Same shell as listing 14.3.2-2.1 on adverse events leading to study drug discontinuation during retreatment phase>>

### Section 14.3.3 – Narratives of deaths, other serious and significant adverse events (non statistics and programming deliverables)

This section does not require statistics and programming deliverables.

#### Section 14.3.4 – Abnormal laboratory value listings

#### Listing 14.3.4-1.1 Listing of abnormal hematology laboratory value – Full Analysis Set

| Country/ Center/<br>Patient/ ARM | Age/ Sex/<br>Race | Phase/ Sample date/<br>Day | Test | Value<br>(SI unit) | Normal<br>range | Grade |
|---|---|---|---|---|---|---|
| XXX/0XXX/0XXXX/X | XX/X/XX | ICONS1/CONS2/TFR/RE-<br>TRT/ DDMMMYYYY/ XX | XXXX | XX (LB/%) | L/N/H | Gx |
| | | ICONS1/CONS2/TFR/RE-<br>TRT/ DDMMMYYYY/ XX | XXXX | XX (LB/%) | L/N/H | Gx |
| XXX/0XXX/0XXXX/X | XX/X/XX | ICONS1/CONS2/TFR/RE-<br>TRT/ DDMMMYYYY/ XX | XXXX | XX (LB/%) | L/N/H | Gx |
| | | ICONS1/CONS2/TFR/RE-<br>TRT/ DDMMMYYYY/ XX | XXXX | XX (LB/%) | L/N/H | Gx |

<sup>-</sup> Arm: 1: Arm 1; 2: Arm 2; 3: Not Randomized.

### Listing 14.3.4-2.1 Listing of abnormal biochemistry laboratory value – Full Analysis Set

<< Programming note: Same shell as listing 14.3.4-1.1 >>

<sup>-</sup> M: Male; F: Female; W: White; B: Black or African American; A: Asian; AI: American Indian or Alaska Native; N: Native Hawaiian or other Pacific Islander; UK: Unknown; O: Other.

<sup>-</sup> Phase: IND = induction phase (0-12 months), CONS1 = pre-randomization consolidation phase (12-24 months), CONS2 = post-randomization consolidation phase (ARM 2)(24-36 months), TFR=treatment free remission phase and RE-TRT=re-treatment phase.

<sup>-</sup> L/H denotes a value below/above normal range, N denotes normal.

<sup>-</sup> Gx denotes an abnormal high value meeting toxicity CTCAE grading criteria and G-x an abnormal low value according to toxicity CTCAE grading. Day is relative to the first day of treatment (day 1).

### **Section 16 – Appendices**

**Section 16.1 – Study information** 

Section 16.1.6 – Listing of patients receiving test drug(s)/investigational product(s) from specific batches where more than one batch was used

Not applicable

Listings (Section 16.1.6)

#### Section 16.1.7 – Randomization scheme and codes (subject identification and treatment assigned)

### Listing 16.1.7-1.1 Randomization schemes - Randomized patients

| Subject ID | Country/<br>Center/<br>Patient | Age/<br>Sex/<br>Race | Randomization<br>date/ Study day | Randomized<br>Treatment | Received<br>Treatment |
|---|---|---|---|---|---|
| | | | DDMMMYYYY/ xx | Arm 1 | Arm 1 |

<sup>-</sup> Randomized patients are all patients meeting eligibility criteria for randomization

<sup>(</sup>i.e. achieved a sustained MR4.0 for at least 12 months in the induction/consolidation phase of the study).

<sup>-</sup> Arm 1: Pre-randomization treatment 24 months, TFR up to 36 months, Re-treatment up to 36 months

<sup>-</sup> Arm 2: Pre-randomization treatment 24 months, Post-randomization treatment 12 months, TFR up to 24 months, Re-treatment up to 24 months.

<sup>-</sup> M: Male; F: Female; W: White; B: Black or African American; A: Asian; AI: American Indian or Alaska Native; N: Native Hawaiian or other Pacific Islander; UK: Unknown; O: Other.

#### **Listings (Section 16.1.7)**

#### Section 16.1.9 – Documentation of statistical methods

This section should include figures, tables and listings for the following data (where applicable):

- inferential analysis outputs for primary & key secondary variables (e.g. additional SAS output)
- any additional information needed about non-inferential analysis outputs

Refer to Guidelines for content of Statistical Appendices of the Clinical Study Report (G029 01)

Guidelines for content of Statistical Appendices of the Clinical Study Report, is available in Cabinets/CREDI TABULU/B&SR/CIS Process Documentation/Guidances (outside of ESOPS)

Attach here shells (a pictorial representation of what the table will look like) or specification (a structured description of a table in words) for each Section 16.1.9 table. Where the layout of a table is exactly the same as a previous table, perhaps with only the population indicator changing, there is no need to repeat the shell each time, simply refer to the previous layout.

Shells may be formatted text or SAS output. Repetition of Section 14 tables is not appropriate.

### Listing 16.1.9.1 Raw Statistical output from Demographic and characteristics at baseline- Full Analysis Set

Insert the contents of the SAS Output Window here.

<<pre><<Pre>rogramming note:

Based on Table 14.1-3.1 Demographic and characteristics at baseline- Full Analysis Set >>

## Listing 16.1.9.1.1 Raw Statistical output from Demographic and characteristics at baseline– LSC sub-study Full Analysis Set

<< Programming note:

Based on Table 14.1-3.1.1 Demographic and characteristics at baseline- LSC sub-study FAS >>

### Listing 16.1.9.2 Raw Statistical output from History of prior Imatinib therapy – Full Analysis Set

<< Programming note:

Based on Table 14.1-5.1 Demographic and characteristics at baseline- Full Analysis Set >>

### Listing 16.1.9.2.1 Raw Statistical output from History of prior Imatinib therapy – LSC sub-study Full Analysis Set

<< Programming note:

Based on Table 14.1-5.1.1 Demographic and characteristics at baseline-LSC sub-study FAS >>

### Listing 16.1.9.3 Raw Statistical output from Cardiovascular risk factors at baseline – Full Analysis Set <<Pre><<Pre><<Pre>rogramming note:

Based on Table 14.1-6.1 Demographic and characteristics at baseline- Full Analysis Set >>

### Listing 16.1.9.4.1 Raw Statistical output from Molecular response MR4.0 at 12 months of TFR-Subset of Full Analysis Set entering the TFR phase

<<Pre>rogramming note:
Based on Table 14.2-2.1.1

### Listing 16.1.9.4.2 Raw Statistical output from Molecular response MR4.0 at 12 months of TFR-Subset of Per Protocol Analysis Set entering the TFR phase

<< Programming note:

Based on Table 14.2-2.1.2 Molecular response MR4.0 at 12 months of TFR-Subset of Per Protocol Set entering the TFR phase >>

### Listing 16.1.9.5.1 Raw Statistical output from Kaplan-Meier analysis of treatment-free survival during the TFR phase – Subset of Full Analysis Set entering the TFR phase

<< Programming note:

Based on Table 14.2-2.2.1 Kaplan-Meier analysis of treatment-free survival during the TFR phase - Subset of Full Analysis Set entering the TFR phase >>

### Listing 16.1.9.5.2 Raw Statistical output from Kaplan-Meier analysis of treatment-free survival during the TFR phase – Subset of Per Protocol Analysis Set entering the TFR phase

<< Programming note:

Based on Table 14.2-2.2.2 Kaplan-Meier analysis of treatment-free survival during the TFR phase - Subset of Per Protocol Analysis Set entering the TFR phase >>

#### Listing 16.1.9.5.3 Raw Statistical output from Kaplan-Meier analysis of overall survival from Randomization– Randomized Set

<< Programming note:

Based on Table 14.2-2.3 Kaplan-Meier analysis of overall survival from Randomization-Randomized Set >>

### Listing 16.1.9.5.4 Raw Statistical output from Kaplan-Meier analysis of progression-free survival during the TFR phase – Subset of Full Analysis Set entering the TFR phase

<< Programming note:

Based on Table 14.2-2.4 Kaplan-Meier analysis of progression-free survival during the TFR phase - Subset of Full Analysis Set entering the TFR phase >>

#### Listing 16.1.9.6.1 Raw Statistical output from Kaplan-Meier estimate of time-to-first CVEs during the prerandomization induction/consolidation phase – Full analysis set

<<pre><<Pre>rogramming note:

Based on Table 14.3.1-11.1.1 Kaplan-Meier analysis of time-to-first CVEs during the pre-randomization induction/consolidation phase - Full analysis set >>

### Listing 16.1.9.6.2 Raw Statistical output from Kaplan-Meier estimate of time-to-first CVEs during the postrandomization consolidation phase (ARM 2)– Subset of Full Analysis Set patients randomized on Arm 2

<< Programming note:

Based on Table 14.3.1-11.1.2 Kaplan-Meier estimate of time-to-first CVEs during the post-randomization consolidation phase (ARM 2) - Subset of Full Analysis Set patients randomized on Arm 2>>

Listing 16.1.9.6.3 Raw Statistical output from Kaplan-Meier estimate of time-to-first CVEs during the retreatment phase – Subset of Full Analysis Set entering the re-treatment phase

<< Programming note:

Based on Table 14.3.1-11.2 Kaplan-Meier estimate of time-to-first CVEs during the re-treatment phase - Subset of Full Analysis Set entering the re-treatment phase >>

RAP Module 7.1 6-May-2021 (14:35) Protocol No CAMN107AIC0

Tables (Section 16.1.9)

### Section 16.2 - Patient data listings

### **Listing 16.2-1.1 Enrolled patients**

| Country/ Center/<br>Patient / ARM | Age/<br>Sex/<br>Race | Date of enrollment | Date of<br>first<br>dose of<br>Nilotinib | Date of last<br>dose of<br>Nilotinib<br>(phase) | Patient entered the re- treatment phase | Date of<br>last<br>contact | Study<br>completion | Study phase<br>discontinuation | Principal cause<br>of phase<br>discontinuation |
|---|---|---|---|---|---|---|---|---|---|
| XXX/0XXX/0XXXX/X<br>XXX/0XXX/0XXXX/X<br>XXX/0XXX/0XXXX/X | XX/X/XX<br>XX/X/XX<br>XX/X/XX | DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY | DDMMMYYYY<br>DDMMMYYYY | DDMMMYYYY/IND<br>DDMMMYYYY/IND<br>DDMMMYYYY/RE-<br>TRT | Yes/No<br>Yes/No<br>Yes/No | DDMMMYYYY<br>DDMMMYYYY | Yes/No<br>Yes/No<br>Yes/No | Yes/No<br>Yes/No<br>Yes/No | XXXXX<br>XXXXX |

<sup>-</sup> Arm: 1: Arm 1; 2: Arm 2; 3: Not Randomized.

<sup>-</sup> M: Male; F: Female; W: White; B: Black or African American; A: Asian; AI: American Indian or Alaska Native; N: Native Hawaiian or other Pacific Islander; UK: Unknown; O: Other.

<sup>-</sup> Phase: IND = induction phase (0-12 months), CONS1 = pre-randomization consolidation phase (12-24 months), CONS2 = post-randomization consolidation phase (ARM 2) (24-36 months), TFR=treatment free remission phase and RE-TRT=re-treatment phase.

<sup>-</sup> Study completion is when EOS visit indicates that study period of 5 years is completed by patient.

<sup>&</sup>lt;< Programming note: For different causes of phase discontinuation use "-" as separator.

### Section 16.2.1 - Discontinued subjects

#### Listing 16.2.1-1.1 Treatment and study completion - Safety Set

| Country/<br>Center/<br>Patient/ Arm | Age/<br>Sex/<br>Race | Last known date on study treatment | Day<br>of last<br>dose | End of study<br>Primary<br>reason # | Followed<br>for survival* | Death<br>Date/Day |
|---|---|---|---|---|---|---|
| | X | 07NOV2005 | 116 | 1 | Yes | 27NOV2005/136 |
| | X | 15SEP2005 | 14 | 2 | Yes | |
| | X | 02MAY2006 | 134 | 7 | No | |
| | X | 16MAR2006 | 17 | 7 | No | |
| | X | 230CT2006 | 119 | 1 | No | |
| | X | 01DEC2006 | 15 | 10 | No | |

<sup>-</sup> Arm: - Arm: 1: Arm 1; 2: Arm 2; 3: Not Randomized. The last known date on study treatment will be taken from DAR page. Day of last dose and Day of death are relative to the first day of treatment (day 1).

# Reason: 1=Adverse event(s), 2=Abnormal laboratory value(s), 3=Abnormal test procedure result(s),
7=Subject withdrew consent, 8=Lost to follow-up, 9=Administrative problems, 10=Death, 16=New cancer (CML) therapy, 17=Disease progression (CML), 25=Protocol deviation, 88=Other, 89=Unstable MR4.0, 90=Pregnancy.

\* Does the subject continue to be followed for survival, stem cell transplantation and disease prog. to AP/BC?
- Patient # reported as disc. Ind/Cons phase due to AE "Blast Crisis" - G2, should have been reported

as disc. Ind/Cons phase due to Disease Progression, progression to Blast Crisis, as per Prot.

### **Listing 16.2.1-1.2 Study discontinuation – Full Analysis Set**

| Phase | Country/ Center/<br>Patient / ARM | Age/ Sex/<br>Race | Date of last<br>dose | Date of end of phase | Reason for discontinuation | Followed for survival |
|---|---|---|---|---|---|---|
| _ | | | | | | |
| CONS1 | | | | | | |
| | XXX/0XXX/0XXXX/2 | XX/X/XX | DDMMMYYYY | DDMMMYYYY | XXXXX | Yes/No |
| | XXX/0XXX/0XXXX/2 | XX/X/XX | DDMMMYYYY | DDMMMYYYY | XXXXX | Yes/No |
| CONS2 | | | | | | |
| | XXX/0XXX/0XXXX/2 | XX/X/XX | DDMMMYYYY | DDMMMYYYY | XXXXX | Yes/No |
| | XXX/0XXX/0XXXX/2 | XX/X/XX | DDMMMYYYY | DDMMMYYYY | XXXXX | Yes/No |
| TFR | | | | | | |
| | XXX/0XXX/0XXXX/X | XX/X/XX | DDMMMYYYY | DDMMMYYYY | XXXXX | Yes/No |
| | XXX/0XXX/0XXXX/X | XX/X/XX | DDMMMYYYY | DDMMMYYYY | XXXXX | Yes/No |
| RE-TRT | | | | | | |
| | XXX/0XXX/0XXXX/X | XX/X/XX | DDMMMYYYY | DDMMMYYYY | XXXXX | Yes/No |
| | XXX/0XXX/0XXXX/X | XX/X/XX | DDMMMYYYY | DDMMMYYYY | XXXXX | Yes/No |

<sup>-</sup> Arm: 1: Arm 1; 2: Arm 2; 3: Not Randomized.

<sup>-</sup> M: Male; F: Female; W: White; B: Black or African American; A: Asian; AI: American Indian or Alaska Native; N: Native Hawaiian or other Pacific Islander; UK: Unknown; O: Other.

<sup>-</sup> Phase: IND = induction phase (0-12 months), CONS1 = pre-randomization consolidation phase (12-24 months), CONS2 = post-randomization consolidation phase (ARM 2)(24-36 months), TFR=treatment free remission phase and RE-TRT=retreatment phase.

<sup>@</sup> For patient # death occurred during Survival follow-up.

<sup>-</sup> Patient reported as disc. Ind/Cons phase due to AE "Blast Crisis"- G2, should have been reported as disc. Ind/Cons phase due to Disease Progression, progression to Blast Crisis, as per Prot.

### Listing 16.2.1-1.3 Screen failures (All subjects enrolled)

| Country/ | Age/ | Date of | _ Criteria not met | | |
|---|---|---|---|---|---|
| Center/<br>Patient | Sex/<br>Race | Screening | Number | Protocol<br>Version | Specific text |
| 0xxxx | | DDMMMYYYY | IC1 | V1 | Male or female patients, aged ≥ 18 years |
| 0xxxx | | DDMMMYYYY | IC3 | V0 | Documented confirmed diagnosis of chronic phase Ph+ and/or BCR-ABL+ CML-CP. |
| 0xxxx | | DDMMMYYYY | IC1 / IC7 | V2 | Male or female patients, aged ≥ 18 years / Patients must have the following electrolyte values within normal limits at screening analysis, or corrected to within normal limits with supplements prior to the first dose of study medication |
| xxxx | | DDMMMYYYY | IC5 / EC3 | V4 | Patient in CCyR (A patient with MMR is considered to be in CCyR / Severe and/or uncontrolled concurrent medical disease |
| • • | | | | | |

<sup>-</sup> M: Male; F: Female;

<sup>-</sup> W: White; B: Black or African American; A: Asian; AI: American Indian or Alaska Native;

N: Native Hawaiian or other Pacific Islander; UK: Unknown; O: Other.

#### Section 16.2.2 - Protocol deviations

### Listing 16.2.2-1.1 Protocol deviations – Enrolled patients

| Country/ Center/<br>Patient/ Arm | Age/ Sex/ Race | Deviation Category | Description of Deviation |
|---|---|---|---|
| XXX/0XXX/0XXXX/X | XX/X/XX | Eligibility/Inclusion | XXXXX |
| XXX/0XXX/0XXXX/X | XX/X/XX | Eligibility/Inclusion | XXXXX |

<sup>-</sup> Arm: 1: Arm 1; 2: Arm 2; 3: Not Randomized.

<sup>-</sup> M: Male; F: Female; W: White; B: Black or African American; A: Asian; AI: American Indian or Alaska Native; N: Native Hawaiian or other Pacific Islander; UK: Unknown; O: Other.

<sup>-</sup> Only major protocol deviation were reported in this listing.

### Section 16.2.3 – Patients excluded from the efficacy analysis

### Listing 16.2.3-1.1 Analysis set - All patients

| Country/ Center/<br>Patient/ Arm | Age/ Sex/<br>Race | Enrolled patients | Full<br>Analysis<br>Set | Randomized<br>Set | Per<br>Protocol<br>Set | Safety<br>Set |
|---|---|---|---|---|---|---|
| XXX/0XXX/0XXXX/X | XX/X/XX | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No |
| XXX/0XXX/0XXXX/X | XX/X/XX | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No |

<sup>-</sup> Arm: 1: Arm 1; 2: Arm 2; 3: Not Randomized.

<sup>-</sup> M: Male; F: Female; W: White; B: Black or African American; A: Asian; AI: American Indian or Alaska Native; N: Native Hawaiian or other Pacific Islander; UK: Unknown; O: Other.

<sup>-</sup> Full Analysis Set (FAS) comprises all subjects who are enrolled, excluding patients with PD severity codes: 0, 8.

<sup>-</sup> Per Protocol Analysis Set (PPS) comprises all subjects who are enrolled without major protocol deviation (PD severity codes: 0, 1, 5, 8).

<sup>-</sup> Safety Set consists of all patients who received at least one dose of study drug, excluding patients with PD severity codes: 0, 5, 8.

### Section 16.2.4 - Demographics and data at screening

### Listing 16.2.4-1.1 Demographic data – Full Analysis Set

| Country/ Center/<br>Patient/ Arm | Age<br>(years) | Sex | If female, child bearing potential* | Race (if other, specify)** | ECOG | BMI | Smoking<br>status | If ex-<br>smoker,<br>duration<br>(months) | <pre>If smoker or ex-smoker, use of tobacco p roduct in the past month***</pre> |
|---|---|---|---|---|---|---|---|---|---|
| XXX/0XXX/0XXXX/X | XX | F/M | XXXXX | XXXXX | 0-5 | XX | No/Yes/Ex | | XXXXX |
| XXX/0XXX/0XXXX/X | XX | F/M | XXXXX | XXXXX | 0-5 | XX | No/Yes/Ex | XX | XXXXX |

<sup>-</sup> Arm: 1: Arm 1; 2: Arm 2; 3: Not Randomized.

### Listing 16.2.4-2.1 Family history – Full Analysis Set

| Country/ Center/<br>Patient/ Arm | Age/ Sex/<br>Race | Diabetes | Hypertension | Dyslipidemia | Cardiac<br>events | Cerebrovascular<br>events | Peripheral<br>arterial<br>disease |
|---|---|---|---|---|---|---|---|
| XXX/0XXX/0XXXX/X | XX/X/XX | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No |
| XXX/0XXX/0XXXX/X | XX/X/XX | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No |

<sup>-</sup> Arm: 1: Arm 1; 2: Arm 2; 3: Not Randomized.

<sup>\*</sup> Able to bear children/ Premenarche/ Post menopausal/ Sterile - of child bearing age.

<sup>\*\*</sup> Caucasian/ Black/ Asian/ Native american/ North african descent/ Unknown/ Other.

<sup>\*\*\*</sup> Cigarettes (including roll-ups/ Cigars/ Tobacco (e.g. pipe)/ Others (e.g. nicotine patches, chewing tobacco).

<sup>-</sup> M: Male; F: Female; W: White; B: Black or African American; A: Asian; AI: American Indian or Alaska Native; N: Native Hawaiian or other Pacific Islander; UK: Unknown; O: Other.

### Listing 16.2.4-2.2 Disease history– Full Analysis Set

| Time from initial diagnosis to screening (months) | Peripheral<br>blood blast<br>at<br>diagnosis<br>(%) | PB | Platelets<br>at<br>diagnosis<br>(10°L) | Spleer<br>size<br>(cm) | Extrame- | Sokal/ Euro (Hasfo rd)/ EUTOS Score (risk) | Molecular<br>response at<br>screening<br>(BCR-ABL(IS)) | Previous progression to AP-BP / Attempt to stop treatment with Imatinib / Have known atypical transcript |
|---|---|---|---|---|---|---|---|---|
| Country: xxx, Age: xxx, Sex xx | | | xxx, arm: | 1/2 | | High/ | | |
| AA | XX | XX | XX | XX | XX | Low/Lo<br>w | >0.01% - <=0.1% | Yes/No/Yes |
| Country: xxx, Age: xxx, Sex xx | | | xxx, arm: | 1/2 | | | | |
| | XX | XX | XX | XX | XX | Low/In<br>termme<br>diate/<br>High | Undetetable | Yes/No/No |

<sup>-</sup> Arm: 1: Arm 1; 2: Arm 2; 3: Not Randomized.

<sup>-</sup> M: Male; F: Female; W: White; B: Black or African American; A: Asian; AI: American Indian or Alaska Native; N: Native Hawaiian or other Pacific Islander; UK: Unknown; O: Other.

<sup>-</sup> Time since initial diagnosis = (date of the baseline visit - date of initial diagnosis)/30.4375.

<sup>-</sup> Extramedullary involvement other than hepato and/or splenomegaly.

<sup>-</sup> Sokal score: low risk (<0.8), intermediate risk (>=0.8-<=1.2) and high risk (>1.2).

<sup>-</sup> Euro (Hasford) score: low risk (<=780), intermediate risk (>780-<=1480) and high risk (>1480).

<sup>-</sup> EUTOS score: low risk (<=87) and high risk (>87).

<sup>-</sup> Molecular response: BCR-ABL (IS): Undetectable; <=0.01%; >0.01% - <=0.1%; >0.1% - <=1%; >1%.

### Listing 16.2.4-3.1 Disease history I– Full Analysis Set

| | | | Diagnosis | | | | |
|---|---|---|---|---|---|---|---|
| Country/<br>Center/<br>Patient/<br>Arm | Age/<br>Sex/<br>Race | Time since initial diagnosis (months) | Peripheral<br>blood<br>blasts % | PB<br>eosinophilis/<br>Basophilis % | Platelets at<br>diagnosis (10E9/L) | Spleen<br>size<br>(cm) | Extramedullary involvement other than hepato and/or splenomegaly |
| XXX/0XXX/0<br>XXXX/X | XX/X/XX | xx.x | XX.X | XX.X | XX.X | XX.X | No |
| XXX/0XXX/0<br>XXXX/X | XX/X/XX | xx.x | XX.X | XX.X | XX.X | XX.X | Yes |

<sup>-</sup> Arm: 1: Arm 1; 2: Arm 2; 3: Not Randomized.

<sup>-</sup> M: Male; F: Female; W: White; B: Black or African American; A: Asian; AI: American Indian or Alaska Native; N: Native Hawaiian or other Pacific Islander; UK: Unknown; O: Other.

#### Listing 16.2.4-3.2 Disease history II– Full Analysis Set

| Country/<br>Center/<br>Patient/<br>Arm | Age/<br>Sex/<br>Race | Time since initial diagnosis (months) | Sokal/<br>Euro<br>(Hasford) /<br>EUTOS<br>score | Sokal<br>score<br>category | Previous<br>progressio<br>n to AP/BC | Attempt to stop<br>treatment<br>with Imatinib | Molecular response<br>at Baseline (BCR-<br>ABL(IS)) |
|---|---|---|---|---|---|---|---|
| XXX/0XXX/0<br>XXXX/X | XX/X/X<br>X | XX.X | xx.x / xx.x / xx.x | low risk | Yes | Yes | >1% |
| XXX/0XXX/0<br>XXXX/X | XX/X/X<br>X | xx.x | xx.x / xx.x / xx.x | intermedia<br>te risk | No | No | Undetectable |

<sup>-</sup> Arm: 1: Arm 1; 2: Arm 2; 3: Not Randomized.

#### Listing 16.2.4-3.3 Medical history/current medical condition – Full Analysis Set

| Country/ Center/<br>Patient/ Arm | Age/ Sex/<br>Race | MedDRA SOC/ Preferred term/ Verbatim | Date of diagnosis/Surgery | Ongoing |
|---|---|---|---|---|
| XXX/0XXX/0XXXX/X | XX/X/XX | SOCXXXXX/PTXXXXX/XXXXX SOCXXXXX/PTXXXXXX | DDMMMYYYY | Yes/No |
| XXX/0XXX/0XXXX/X | XX/X/XX | | DDMMMYYYY | Yes/No |

<sup>-</sup> Arm: 1: Arm 1; 2: Arm 2; 3: Not Randomized.

<sup>-</sup> M: Male; F: Female; W: White; B: Black or African American; A: Asian; AI: American Indian or Alaska Native; N: Native Hawaiian or other Pacific Islander; UK: Unknown; O: Other.

<sup>-</sup> Sokal score: low risk (<0.8), intermediate risk (>=0.8-<=1.2) and high risk (>1.2).

<sup>-</sup> Baseline is defined as the last available assessment before or at date of start of study treatment.

<sup>-</sup> Molecular response: BCR-ABL (IS): Undetectable; <=0.01%; >0.01% - <=0.1%; >0.1% - <=1%; >1%.

<sup>-</sup> M: Male; F: Female; W: White; B: Black or African American; A: Asian; AI: American Indian or Alaska Native; N: Native Hawaiian or other Pacific Islander; UK: Unknown; O: Other.
RAP Module 7.1 6-May-2021 (14:35) Protocol No CAMN107AIC0

# Listing 16.2.4.4 Cardiovascular risk factors at baseline for patients with not evaluable CV risk factor, Full Analysis Set

| CVEs<br>history | Diabetes<br>mellitus<br>history | Hypertension<br>history | Severe<br>hypertension<br>history | Dyslipidemia<br>history | Familial<br>dyslipidemia<br>history | Systolic<br>blood<br>pressure<br>(mmHg) | Total<br>cholesterol<br>(mmol/L) | Micro-<br>albuminuria<br>(mg/L) | Creatinine<br>(umol/L) | G<br>F<br>R | Heart<br>score |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Country: xxx,<br>Smoking status<br>Date of first | s: xxx, Wei | ght (kg): xxx | , BMI (kg/m2) | • | e: xxx | | | | | | |
| Yes (IHD/<br>PAOD/ ICE/<br>OTHER) /No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | XX | XX | XX | XX | X<br>X | XX |

<sup>-</sup> Arm: 1: Arm 1; 2: Arm 2; 3: Not Randomized.

GFR = [(140-age)\*weight (kg)\*0.85 (for women)] / [Cr (umol/1)\*0.814].

#### << Programming note:

Date of first study medication: STTEXP10 [derived.a\_ dar]

CVEs history: CVEMH [derived.a ident]

Diabetes mellitus history: CVDBTMH [derived.a\_ ident]

Hypertension history: CVHYPMH [derived.a ident]

Severe hypertension history: CVSEHYMH [derived.a ident]

Dyslipidemia history: CVDYSMH [derived.a\_ ident]

Familial dyslipidemia history: CVFADYMH [derived.a ident]

Systolic Blood pressure: STNSBPB [derived.a ident]

Total cholesterol: TCHOLB [derived.a\_ ident] Micro-albuminuria : UMALBB [derived.a\_ ident]

Creatinine: CREATB [derived.a ident]

GFR: CVGFR [derived.a ident]

Heart Score: HSCORE [derived.a ident] >>

<sup>-</sup> IHD: Ischemic heart disease, PAOD: Peripheral arterial occlusive disease, ICE: Ischemic cerebrovascular events.

<sup>-</sup> GFR measured by Cockcroft-Gault Creatinine Clearance rate as defined below:

<sup>-</sup> HeartScore defined by the European Guidelines on cardiovascular disease prevention in clinical practice (version 2012) and based on age, gender, smoking status, systolic blood pressure, total cholesterol and country.

### Section 16.2.5 – Compliance and/or drug concentration data if available (including Bioanalytical Data Report)

### Listing 16.2.5-1.1 Dosage administration records – Full Analysis Set

| Country/ Center/<br>Patient/ Arm | Age/ Sex/<br>Race | Drug administration<br>Start/End dates | Phase | Total Dose<br>(mg/day)/ Frequency | Discontinuation* | Reason for<br>Discontinuation |
|---|---|---|---|---|---|---|
| XXX/0XXX/0XXXX/X | XX/X/XX | DDMMMYYYY/ DDMMMYYYY | IND/CONS | XX/XX | | _ |
| XXX/0XXX/0XXXX/X | XX/X/XX | DDMMMYYYY/ DDMMMYYYY | TFR | XX/XX | | |
| XXX/0XXX/0XXXX/X | XX/X/XX | DDMMMYYYY/ DDMMMYYYY | RE-TRT | XX/XX | XXXXX | XXXXX |

<sup>-</sup> Arm: 1: Arm 1; 2: Arm 2; 3: Not Randomized.

### Section 16.2.6 – Individual efficacy response data

# Listing 16.2.6-1.1 BCR-ABL(IS) ratio and molecular responses during Induction/Consolidation and post-randomization consolidation phase (ARM 2) – Full Analysis Set

| Country/ Center/<br>Patient/ Arm | Age/ Sex/ Race Vi | .sit Time-<br>window/Day | BCR-ABL(IS) ratio (%) | Total number of ABL copies | Molecular response |
|---|---|---|---|---|---|
| XXX/0XXX/0XXXX/X | XX/X/XX | | | | |
| | Ba | aseline | XX | XX | MMR/MR4.0/MR4.5 |
| | 31 | 1 | XX | XX | MMR/MR4.0/MR4.5 |
| | Repeat | t at each time-point ev | ery 3 month ti | 11 24/36 months | |
| XXX/0XXX/0XXXX/X | XX/X/XX | | | | |
| | Ba | aseline | XX | XX | MMR/MR4.0/MR4.5 |
| | 31 | 1 | XX | XX | MMR/MR4.0/MR4.5 |
| | Repeat | t at each time-point ev | ery 3 month ti | 11 24/36 months | |

<sup>-</sup> Arm: 1: Arm 1; 2: Arm 2; 3: Not Randomized.

<sup>\*</sup> Discontinuation: None/Changed/Interrupted/Permanently.

<sup>-</sup> Phase: IND/CONS = induction/consolidation phase, TFR=treatment free remission phase and RE-TRT=re-treatment phase.

<sup>-</sup> M: Male; F: Female; W: White; B: Black or African American; A: Asian; AI: American Indian or Alaska Native; N: Native Hawaiian or other Pacific Islander; UK: Unknown; O: Other.

<sup>-</sup> Patient # reported as disc. Ind/Cons phase due to AE "Blast Crisis"- G2, should have been reported as disc. Ind/Cons phase due to Disease Progression, progression to Blast Crisis, as per Prot.

<sup>-</sup> M: Male; F: Female; W: White; B: Black or African American; A: Asian; AI: American Indian or Alaska Native; N: Native Hawaiian or other Pacific Islander; UK: Unknown; O: Other.

- Patients randomized to Arm 1 have 24 months of treatment and a maximum of 36 months of re-treatment.
- Patients randomized to Arm 2 have 36 months of treatment and a maximum of 24 months of re-treatment.

## Listing 16.2.6-1.2 BCR-ABL(IS) ratio and molecular responses during TFR phase – Subset of Full Analysis Set entering the TFR phase

| Country/ Center/<br>Patient/ Arm | Age/ Sex/ Race | (/igit | Time-<br>window/Day | BCR-ABL(IS) ratio (%) | Total number of ABL copies | Molecular response |
|---|---|---|---|---|---|---|
| XXX/0XXX/0XXXX/X | XX/X/XX | | | | | |
| | ] | Baseline | | XX | XX | MMR/MR4.0/MR4.5 |
| | : | 3M | | XX | XX | MMR/MR4.0/MR4.5 |
| XXX/0XXX/0XXXX/X | Repeat at each tin<br>XX/X/XX | me-point every | / 3 month ti | ll 24/36 mont | hs | |
| | ] | Baseline | | XX | XX | MMR/MR4.0/MR4.5 |
| | : | 3M | | XX | XX | MMR/MR4.0/MR4.5 |
| | Repeat at each ti | me-point every | / 3 month ti. | ll 24/36 mont | hs | |

<sup>-</sup> Arm: 1: Arm 1; 2: Arm 2; 3: Not Randomized.

# Listing 16.2.6-1.3 BCR-ABL(IS) ratio and molecular responses during re-treatment phase – Subset of Full Analysis Set entering the re-treatment phase

<< Same shell as listing 16.2.6-1.2 with the following second footnote:

- Patients randomized to Arm 1 have 24 months of treatment and a maximum of 36 months of re-treatment.
- Patients randomized to Arm 2 have 36 months of treatment and a maximum of 24 months of re-treatment. >>

<sup>-</sup> M: Male; F: Female; W: White; B: Black or African American; A: Asian; AI: American Indian or Alaska Native; N: Native Hawaiian or other Pacific Islander; UK: Unknown; O: Other.

<sup>-</sup> Patients randomized to Arm 1 have a miximum of 36 months of TFR phase;

<sup>-</sup> Patients randomized to Arm 2 have a maximum of 24 months of TFR phase;

### Listing 16.2.6-2.1 Criteria of successful TFR – Subset of Full Analysis Set entering the TFR phase

| Country/ Center/<br>Patient/ Arm | Age/<br>Sex/<br>Race | Visit | Time-window/<br>Day | Loss of<br>MMR | Loss of MR4.0 | Confirmed loss of MR4.0 | Re-start of<br>Nilotinib | Successful<br>TFR at<br>Month 12 |
|---|---|---|---|---|---|---|---|---|
| XXX/0XXX/0XXXX/X | XX/X/XX | V101-A1-Month 1 | M1/35 | Yes/No | Yes/No | Yes/No | Yes/No | |
| | | V106-A1-Month 6 | M6/190 | Yes/No | Yes/No | Yes/No | Yes/No | |
| | | | Repeat at all | TFR visits | | | | |
| | | V109-A1-Month 12 | M12/408 | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No |
| | | V401-EOP-TFR | M12/420 | Yes/No | Yes/No | Yes/No | Yes/No | |
| XXX/0XXX/0XXXX/X | XX/X/XX | | м3/90 | Yes/No | Yes/No | Yes/No | Yes/No | |
| | | | M6/190 | Yes/No | Yes/No | Yes/No | Yes/No | |
| | | | Repeat at all | TFR visits | | | | |

<sup>-</sup> Arm: 1: Arm 1; 2: Arm 2; 3: Not Randomized.

<sup>\*</sup> in case of unsuccessful TFR, put 'No' on the row with confirmed loss of MR4.0=Yes or re-start of nilotinib=Yes.

<sup>-</sup> M: Male; F: Female; W: White; B: Black or African American; A: Asian; AI: American Indian or Alaska Native; N: Native Hawaiian or other Pacific Islander; UK: Unknown; O: Other.

<sup>-</sup> Confirmed loss of MR4.0 defined as three consecutive tests less than MR4.0 assessed at three consecutive visits.

<sup>-</sup> Successful TFR is defined as MR4.0, no confirmed loss of MR4.0, no loss of MMR and no re-starting of nilotinib therapy at the end of 12 months in the TFR phase of the study.

<sup>-</sup> Patients randomized to Arm 1 have a maximum of 36 months of TFR phase; Patients randomized to Arm 2 have a maximum of 24 months of TFR phase;

# Listing 16.2.6-3.1 Assessment of progression-free survival during the TFR phase –Subset of Full Analysis Set entering the TFR phase

| Country/ Center/<br>Patient/Arm | Age/ Sex/<br>Race | Progression | Date of progression | Time to progression/censoring (months) | Type of progression |
|---|---|---|---|---|---|
| XXX/0XXX/0XXXX\X | XX/X/XX | Yes/No | DDMMMYYYY | XX | XXXXX |
| XXX/0XXX/0XXXX\X | XX/X/XX | Yes/No | DDMMMYYYY | XX | XXXXX |

<sup>-</sup> Arm: 1: Arm 1; 2: Arm 2; 3: Not Randomized.

Censoring rule = patients who did not meet the event are censored at the first date occurring between: the last contact date, the end of TFR phase, the DBL date and the date of death.

<sup>-</sup> M: Male; F: Female; W: White; B: Black or African American; A: Asian; AI: American Indian or Alaska Native; N: Native Hawaiian or other Pacific Islander; UK: Unknown; O: Other.

<sup>-</sup> Event = first occurrence of progression to AP/BC or death for any cause.

<sup>-</sup> Time to event = (date of event - start date of TFR phase + 1)/30.4375.

<sup>-</sup> Patients randomized to Arm 1 have a miximum of 36 months of TFR phase; Patients randomized to Arm 2 have a maximum of 24 months of TFR phase.

# Listing 16.2.6-3.2 Assessment of treatment-free survival during the TFR phase –Subset of Full Analysis Set entering the TFR phase

| Country/ Center/<br>Patient/Arm | Age/ Sex/<br>Race | Treatment free | Date of event | Time from Day 1 of<br>TFR to<br>event/censoring<br>(months) | Type of event |
|---|---|---|---|---|---|
| XXX/0XXX/0XXXX\X | XX/X/XX | Yes/No | DDMMMYYYY | XX | XXXXX |
| XXX/0XXX/0XXXX\X | XX/X/XX | Yes/No | DDMMMYYYY | XX | XXXXX |

<sup>-</sup> Arm: 1: Arm 1; 2: Arm 2; 3: Not Randomized.

<sup>-</sup> M: Male; F: Female; W: White; B: Black or African American; A: Asian; AI: American Indian or Alaska Native; N: Native Hawaiian or other Pacific Islander; UK: Unknown; O: Other.

<sup>-</sup> Event = first occurrence of relapse, re-treatment with nilotinib, progression to AP/BC or death for any cause. Censoring rule = patients who did not meet the event are censored at the first date occurring between: the last contact date, the end of TFR phase, the DBL date and the date of death.

<sup>-</sup> Time to event = (date of event - start date of TFR phase + 1)/30.4375.

<sup>-</sup> Patients randomized to Arm 1 have a miximum of 36 months of TFR phase; Patients randomized to Arm 2 have a maximum of 24 months of TFR phase.

### Listing 16.2.6-3.3 Assessment of overall survival From Randomization – Randomized set

| Country/ Center/<br>Patient/Arm | Age/ Sex/<br>Race | Alive | Date of event(death) | Time from Randomization to death /censoring (months) |
|---|---|---|---|---|
| XXX/0XXX/0XXXX\X | XX/X/XX | Yes/No | DDMMMYYYY | XX |
| XXX/0XXX/0XXXX\X | XX/X/XX | Yes/No | DDMMMYYYY | XX |

<sup>-</sup> Arm: 1: Arm 1; 2: Arm 2; 3: Not Randomized.

Censoring rule = patients who did not meet the event are censored at the first date occurring between: the last contact date, and the date of death.

<sup>-</sup> M: Male; F: Female; W: White; B: Black or African American; A: Asian; AI: American Indian or Alaska Native; N: Native Hawaiian or other Pacific Islander; UK: Unknown; O: Other.

<sup>-</sup> Event = death for any cause.

<sup>-</sup> Time to event = (date of event - Randomization date + 1)/30.4375.

# Listing 16.2.6-3.4 Assessment of relapse and treatment status during the TFR phase –Subset of Full Analysis Set entering the TFR phase and relapsed

| | | | | | Start of re-tr | reatment after Relapse |
|---|---|---|---|---|---|---|
| Country/ Center/<br>Patient/Arm | Age/<br>Sex/<br>Race | Date of<br>Relapse | Time from Day 1 of TFR to relapse (months) | Re-treatment | Date | Days after relapse. |
| XXX/0XXX/0XXXX\X | XX/X/XX | DDMMMYYYY | XX | Yes | DDMMMYYYY | XX |
| XXX/0XXX/0XXXX\X | XX/X/XX | DDMMMYYYY | XX | No | | |

<sup>-</sup> Arm: 1: Arm 1; 2: Arm 2; 3: Not Randomized.

<sup>-</sup> M: Male; F: Female; W: White; B: Black or African American; A: Asian; AI: American Indian or Alaska Native; N: Native Hawaiian or other Pacific Islander; UK: Unknown; O: Other.

<sup>-</sup> Time to event = (date of relapse - start date of TFR phase + 1)/30.4375.

<sup>-</sup> Patients randomized to Arm 1 have a maximum of 36 months of TFR phase; Patients randomized to Arm 2 have a maximum of 24 months of TFR phase;

# Listing 16.2.6-4.1 WBC and molecular response in patients with WBC increase (CTCAE grade>G1) – Full Analysis Set

| Country/<br>Center/<br>Patient/Arm | Age/<br>Sex/<br>Race/ | Time-<br>point | Visit | Lab sample<br>date/day | WBC<br>10E9/L | RQ-PCR sample<br>date/day | Molecul<br><u>Respon</u><br>eCRF De | se |
|---|---|---|---|---|---|---|---|---|
| | /x | M3 | V1-M3 | xxxxxxxx/98 | xxx Gx | xxxxxxxx/98 | MMR MI | MR |
| | | М6 | V2-M6 | | | xxxxxxxxx/183 | MR4.0 M | R4.0 |
| | | М6 | UNSCH | xxxxxxxx/186 | xxx Gx | | | |
| | /x | XX | xxxxx | xxxxxxxx/xxx | xxx Gx | xxxxxxxx/xxx | xxxx x | xxx |
| | | XX | XXXXX | xxxxxxxx/xxx | xxx Gx | xxxxxxx/xxx | XXXX X | XXX |
| | | XX | XXXXX | xxxxxxxx/xxx | xxx Gx | xxxxxxx/xxx | XXXX X | XXX |
| | - | XX | XXXXX | xxxxxxxx/xxx | xxx Gx | xxxxxxxx/xxx | XXXX X | xxx |

<sup>-</sup> Arm: 1: Arm 1; 2: Arm 2; 3: Not Randomized.

<< Programming note: For each patient merge PCR data with haematological data by time-point and visit. If there are several unscheduled visit in a time-window then merge them by incremental order defined by chronology >>;

<sup>-</sup> Gx denotes a value meeting toxicity grading criteria (NCI-CTCAE version 4.03).

<sup>-</sup> Note: EOP = End Of Phase; UNSCH = Unscheduled visit.

## Listing 16.2.6-5.1 Individual Efficacy data, Molecular response – Full Analysis Set

| | | | | | | | | | Molecu<br>Respon | |
|---|---|---|---|---|---|---|---|---|---|---|
| Country/<br>Center/<br>Patient/Arm | Age/<br>Sex/<br>Race | Time-<br>point | Visit | Evaluation<br>was not<br>done | RQ-PCR<br>sample<br>date/day | Evaluation not evaluable | Total<br>ABL<br>copies | BCR-<br>ABL<br>(IS)<br>(%) | eCRF | Derived |
| | | • | | | | | | | | |
| /x | | М3 | V1-M3 | | xxxxxxxxx/98 | | XXXXXX | XX.X | 3 | 3 |
| | | М6 | V2-M6 | N.D. | | | | | | |
| | | | | | | N.E. | | | | |
| /x | | MX | VX-MX | | xxxxxxxxx/XX | | xxxxxx | XX.X | 3 | 3 |
| / 25 | | MX | VX-MX | | xxxxxxxxx/XX | | XXXXXX | XX.X | 4.0 | 4.0 |
| | | | | | | | ••• | | | |
| | | <b></b> | | | | | | | | |
| /x | | MX | VX-MX | | xxxxxxxx/XX | | xxxxx | XX.X | 4.0 | 3.0 |
| | | MX | VX-MX | | xxxxxxxxx/XX | | XXXXXX | XX.X | 5.0 | 4.5 |
| | | ••• | | | | | | | ••• | |
| ••• | | *** | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• |

<sup>-</sup> Arm: 1: Arm 1; 2: Arm 2; 3: Not Randomized.

<sup>-</sup> Note: EOP = End Of Phase; UNSCH = Unscheduled visit, N.D.: Not Done, N.E.: Not evaluable.

## Listing 16.2.6-5.2 Individual Efficacy data, Bone-marrow I – Full Analysis Set

| | | | | | | | | | Pero | cent of | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Country/<br>Center/<br>Patient/Arm | Age/<br>Sex/<br>Race | Time-<br>point | Visit | Evaluat<br>ion was<br>not<br>done | Bone-arrow<br>sample<br>date/day | Bone marrow sample collected | Cellularity | Blasts | Pro<br>Myelo-<br>cytes | Baso-<br>philis | Eosino-<br>philis |
| | | мз | V1-M3 | | xxxxxxxxx/98 | Aspirate | Hypocellular | XX.X | XX.X | XX.X | XX.X |
| | | М6 | V2-M6 | N.D. | | | | | | | |
| | | MX | VX-MX | | xxxxxxxxx/XX | Aspirate | Normocellular | XX.X | XX.X | XX.X | XX.X |
| | | MX | VX-MX | | xxxxxxxxx/XX | Aspirate | Hypocellular | XX.X | xx.x | XX.X | XX.X |
| | | | | | | - | | | | | |
| | | MX | VX-MX | | xxxxxxxx/XX | Biopsy | Normocellular | XX.X | XX.X | XX.X | XX.X |
| | | MX | VX-MX | | xxxxxxxxx/XX | Aspirate | Hypocellular | xx.x | xx.x | XX.X | xx.x |
| | | ••• | | | | - | - | | ••• | | |
| | | ••• | | ••• | | | | | ••• | ••• | |

<sup>-</sup> Arm: 1: Arm 1; 2: Arm 2; 3: Not Randomized.

<sup>-</sup> Note: EOP = End Of Phase; UNSCH = Unscheduled visit, N.D.: Not Done.

## Listing 16.2.6-5.3 Individual Efficacy data, Bone -marrow II – Full Analysis Set

| | | | | | | | Number of metaphases | | ases | Additional aberrations | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Country/<br>Center/<br>Patient/Arm | Age/<br>Sex/<br>Race | Time-<br>point | Visit | Evaluat<br>ion was<br>not<br>done | Bone-arrow<br>sample<br>date/day | Bone marrow sample collected | Analyzed | Ph + | Ph - | Ph + | Ph - |
| | | мз | V1-M3 | | xxxxxxxxx/98 | Aspirate | XXX | XXX | XXX | Yes | No |
| /x | | М6 | V2-M6 | | xxxxxxxxx/186 | Biopsy | XXX | XXX | xxx | No | No |
| | | | | | | 1 - 2 | | | | | |
| | | | | | / | | | | | | |
| \x | | MX | VX-MX | | xxxxxxxx/XX | Aspirate | XXX | XXX | XXX | No | Yes |
| | | MX | VX-MX | N.D. | | | | | | | |
| | | | | | | | | | | ••• | |
| | | MX | VX-MX | | xxxxxxxx/XX | Biopsy | xxx | xxx | xxx | No | No |
| /x | | | | | | | | | | | |
| | | MX<br> | VX-MX<br> | | xxxxxxxx/XX<br> | Aspirate | XXX | XXX<br> | xxx<br> | Yes<br> | Yes<br> |
| | | ••• | ••• | | | | | ••• | | ••• | |
| | | | ••• | ••• | | | ••• | | ••• | | ••• |

<sup>-</sup> Arm: 1: Arm 1; 2: Arm 2; 3: Not Randomized.

<sup>-</sup> Note: EOP = End Of Phase; UNSCH = Unscheduled visit, N.D.: Not Done.

### Listing 16.2.6-6.1.1 Total percentage of CD34+ cells – LSC sub-study Full Analysis Set

| Country/ Center/ Patient/ Arm | Age/ Sex/ Race | Time point | Total CD34+ |
|-------------------------------|----------------|------------|-------------|
| XXX/0XXX/0XXXX/X | XX/X/XX | Screening# | XXX.X |
| XXX/0XXX/0XXXX/X | XX/X/XX | Month 24 | XXX.X |
| XXX/0XXX/0XXXX/X | XX/X/XX | Month 36 | XXX.X |
| XXX/0XXX/0XXXX/X | XX/X/XX | EOP TFR | XXX.X |

<sup>-</sup> Arm: 1: Arm 1; 2: Arm 2; 3: Not Randomized.

<sup>-</sup> M: Male; F: Female; W: White; B: Black or African American; A: Asian; AI: American Indian or Alaska Native;

N: Native Hawaiian or other Pacific Islander; UK: Unknown; O: Other.

<sup>#</sup> Baseline value, latest available valid evaluation between Screening and Rescreening.

### Listing 16.2.6-6.2.1 Percentage of cells from total CD34 positive— LSC sub-study Full Analysis Set

Percentage from total CD34+

| Country/ Center/<br>Patient/ Arm | Age/<br>Sex/<br>Race | Time<br>point | CD34+/CD38+ | CD34+/CD38- | Immunopheno-<br>typically<br>Aberrant<br>CD34+ cells | Immunopheno-<br>typically<br>Aberrant CD34<br>Negative cells |
|---|---|---|---|---|---|---|
| XXX/0XXX/0XXXX/X | XX/X/XX | Screening# | XXX.X | XXX.X | XXX.X | XXX.X |
| | | Month 24 | XXX.X | XXX.X | XXX.X | XXX.X |
| | | Month 36 | XXX.X | XXX.X | XXX.X | XXX.X |
| | | EOP TFR | XXX.X | XXX.X | XXX.X | XXX.X |
| XXX/0XXX/0XXXX/X | XX/X/XX | Screening | XXX.X | XXX.X | XXX.X | XXX.X |
| | | Re-screening# | XXX.X | XXX.X | XXX.X | XXX.X |
| | | Month 24 | XXX.X | XXX.X | XXX.X | XXX.X |
| | | Month 36 | XXX.X | XXX.X | XXX.X | XXX.X |
| | | EOP TFR | XXX.X | XXX.X | XXX.X | XXX.X |

<sup>-</sup> Arm: 1: Arm 1; 2: Arm 2; 3: Not Randomized.

<sup>-</sup> M: Male; F: Female; W: White; B: Black or African American; A: Asian; AI: American Indian or Alaska Native;

N: Native Hawaiian or other Pacific Islander; UK: Unknown; O: Other.

<sup>#</sup> Baseline value, latest available valid evaluation between Screening and Rescreening.

### Listing 16.2.6-6.3.1 Number of events sorted- LSC sub-study Full Analysis Set

| Country/ Center/<br>Patient/ Arm | Age/<br>Sex/<br>Race | Time<br>point | CD34+/CD38+ | CD34+/CD38- | Immunopheno-<br>typically<br>Aberrant<br>CD34+ cells | Immunopheno-<br>typically<br>Aberrant CD34<br>negative cells |
|---|---|---|---|---|---|---|
| XXX/0XXX/0XXXX/X | XX/X/XX | Screening# | XXX.X | XXX.X | XXX.X | XXX.X |
| | | Month 24 | XXX.X | XXX.X | XXX.X | XXX.X |
| | | Month 36 | XXX.X | XXX.X | XXX.X | XXX.X |
| | | EOP TFR | XXX.X | XXX.X | XXX.X | XXX.X |
| XXX/0XXX/0XXXX/X | XX/X/XX | Screening | XXX.X | XXX.X | XXX.X | XXX.X |
| | | Re-screening# | XXX.X | XXX.X | XXX.X | XXX.X |
| | | Month 24 | XXX.X | XXX.X | XXX.X | XXX.X |
| | | Month 36 | XXX.X | XXX.X | XXX.X | XXX.X |
| | | EOP TFR | XXX.X | XXX.X | XXX.X | XXX.X |

<sup>-</sup> Arm: 1: Arm 1; 2: Arm 2; 3: Not Randomized.

<sup>-</sup> M: Male; F: Female; W: White; B: Black or African American; A: Asian; AI: American Indian or Alaska Native; N: Native Hawaiian or other Pacific Islander; UK: Unknown; O: Other.

<sup>#</sup> Baseline value, latest available valid evaluation between Screening and Rescreening.

Immunopheno-

Immunopheno-

## Listing 16.2.6-6.4.1 Ph+ by HIS- LSC sub-study Full Analysis Set

| Country/ Center/<br>Patient/ Arm | Age/<br>Sex/<br>Race | Time<br>point | CD34+/CD38+<br>(Percentage<br>of Ph+) | CD34+/CD38-<br>(Percentage of<br>Ph+) | typically Aberrant CD34+ cells (Percentage of Ph+) | typically<br>aberrant CD34<br>negative<br>cells<br>(Percentage<br>of Ph+) |
|---|---|---|---|---|---|---|
| XXX/0XXX/0XXXX/X | XX/X/XX | Screening# | Positive (xx.x%) | Negative | Missing | Missing |
| | | Month 24 | Positive (xx.x%) | Negative | Positive (xx.x%) | Positive (xx.x%) |
| | | Month 36 | Positive (xx.x%) | Negative | Negative | Negative |
| | | EOP TFR | XXX.X | XXX.X | XXX.X | XXX.X |
| XXX/0XXX/0XXXX/X | XX/X/XX | Screening | Negative | Not Evaluable | Positive (xx.x%) | Positive (xx.x%) |
| | | Re-screening# | Negative | Not Evaluable | Positive (xx.x%) | Positive (xx.x%) |
| | | Month 24 | Positive (xx.x%) | Negative | Negative | Negative |
| | | Month 36 | Positive (xx.x%) | Positive (xx.x%) | Negative | Negative |
| | | EOP TFR | XXX.X | XXX.X | XXX.X | XXX.X |

<sup>-</sup> Arm: 1: Arm 1; 2: Arm 2; 3: Not Randomized.

<sup>-</sup> M: Male; F: Female; W: White; B: Black or African American; A: Asian; AI: American Indian or Alaska Native; N: Native Hawaiian or other Pacific Islander; UK: Unknown; O: Other.

<sup>#</sup> Baseline value, latest available valid evaluation between Screening and Rescreening.

## Listing 16.2.6-6.5.1 BCR-ABL by RT-PCR- LSC sub-study Full Analysis Set

| Country/ Center/<br>Patient/ Arm | Age/<br>Sex/<br>Race | Time<br>point | CD34+/CD38+ | CD34+/CD38- | Immunopheno-<br>typically<br>Aberrant<br>CD34+ cells | Immunopheno-<br>typically<br>aberrant CD34<br>negative<br>cells |
|---|---|---|---|---|---|---|
| XXX/0XXX/0XXXX/X | XX/X/XX | Screening# | Positive | Negative | Missing | Missing |
| | | Month 24 | Positive | Negative | Positive | Positive |
| | | Month 36 | Positive | Negative | Negative | Negative |
| | | EOP TFR | XXX.X | XXX.X | XXX.X | XXX.X |
| XXX/0XXX/0XXXX/X | XX/X/XX | Screening | Negative | Not Evaluable | Positive | Positive |
| | | Re-screening# | Negative | Not Evaluable | Positive | Positive |
| | | Month 24 | Positive | Negative | Negative | Negative |
| | | Month 36 | Positive | Positive | Negative | Negative |
| | | EOP TFR | XXX.X | XXX.X | XXX.X | XXX.X |

<sup>-</sup> Arm: 1: Arm 1; 2: Arm 2; 3: Not Randomized.

<sup>-</sup> M: Male; F: Female; W: White; B: Black or African American; A: Asian; AI: American Indian or Alaska Native; N: Native Hawaiian or other Pacific Islander; UK: Unknown; O: Other.

<sup>#</sup> Baseline value, latest available valid evaluation between Screening and Rescreening.

### Section 16.2.7 – Adverse event listings

### Listing 16.2.7-1.1 All adverse events – Full Analysis Set

| Country/ Center/<br>Patient/ Arm | Age/ Sex/<br>Race | Adverse Event Verbatim/<br>Abbreviated System organ<br>class/ Preferred term | Start<br>date/day | End<br>date/day | Dur.<br>(days) | Phase | Grade/SAE/ Relation/<br>Action taken |
|---|---|---|---|---|---|---|---|
| XXX/0XXX/0XXXX/X | XX/X/XX | XXXXX/SOCXXXXX/PTXXXXX | DDMMMYYYY/X^ | DDMMMYYYY/X | XX | IND/CON<br>S | G0-5/No/NS-S/A0-5 |
| XXX/0XXX/0XXXX/X | XX/X/XX | XXXXX/SOCXXXXX/PTXXXXX | DDMMMYYYY/X^ | DDMMMYYYY/X | XX | TFR | G0-5/Yes/NS-S/A0-5 |
| XXX/0XXX/0XXXX/X | XX/X/XX | XXXXX/SOCXXXXX/PTXXXXX | DDMMMYYYY/X* | DDMMMYYYY/X | XX | RE-TRT | G0-5/No/NS-S/A0-5 |

- Arm: 1: Arm 1; 2: Arm 2; 3: Not Randomized.- M: Male; F: Female; W: White; B: Black or African American; A: Asian; AI: American Indian or Alaska Native; N: Nat. Hawaiian or other Pac. Isl.; UK: Unknown; O: Other. Day is relative to the first day of Treat. (day 1). Relationship to study drug: NS=Not suspected, S=Suspected.
- Action taken: A0=No action taken; A1=Study drug dosage adj./temp. inter.; A2=Study drug perm. Discount. due to this AE; A3=Concomitant med. taken; A4=Non-drug therapy given; A5=Hosp./Prolonged hosp.

Phase: IND/CONS = ind./Cons. phase, TFR=treat. free remission phase and RE-TRT=re-treat. phase.

- \* Event occurred more than 30 days after last study treatment exposure date.
- ^ Event occurred between patient's informed consent date and the day before first dose of study medication.
- @ For patient # death occurred during Survival follow-up.

<<Pre>rogramming note: Abbreviated system organ class to be used for the listings i.e. removing the term disorder and
conditions:

"NEOPLASMS"; "RESPIRATORY"; "BLOOD"; "GI"; "GENERAL"; "INFECTIONS"; "INJURIES"; "MUSCULOSKELETAL"; "NERVOUS"; "RENAL"; "REPRODUCTIVE SYSTEM"; "SKIN"; "SURGICAL AND MEDICAL"; "METABOLISM"; "IMMUNE".>>

#### Add the following text in the main body of the Listing's last page:

- Patient reported as disc. Ind/Cons phase due to AE "Blast Crisis" G2, should have been reported as disc. Ind/Cons phase due to Disease Progression, progression to Blast Crisis, as per Prot.
- For patient # AE "PHLEGMON FOOT BIG TOE RIGHT" is reported as PT "Cellulitis" in the AE listing while it is reported as PT "Osteoarthritis" in the SAE listing. PT for the same AE has been wrongly decoded and reconciliation was not requiring a perfect match of the PT.

#### Add following footnote at the end of last page:

- For patient # \_\_\_\_\_, due to reconciliation discrepancies, safety database reported AE term "Endometriosis" as a SAE, while in clinical database this AE was not recorded as an SAE.

### Listing 16.2.7-2.1 Serious adverse events Full Analysis Set

| Country/<br>Center/<br>Patient/<br>Arm | | Age/<br>Sex/<br>Race | Adverse Event Verbatim/<br>Abbreviated System organ<br>Preferred term | class/ | Start<br>date/<br>day | End<br>date/<br>day | Duration<br>(days) | Gradfe/<br>Relation/<br>Action<br>taken |
|---|---|---|---|---|---|---|---|---|
| | /x | | Verbatim/Ab SOCxxxxxx<br>Verbatim/Ab SOCxxxxxx | , | 16JUL2005/2<br>18JUL2005/4* | 27JUL2005/13<br>27JUL2005/13 | | G1/NS/A0<br>G1/S/A3,5 |

16JUL2005/-1^ 27JUL2005/13 12

G1/NS/A0

Verbatim/Ab SOCxxxxxx / PTxxxxxxxxxxx

<< Programming note: Abbreviated system organ class to be used for the listings i.e. removing the term disorder and conditions:

"NEOPLASMS"; "RESPIRATORY"; "BLOOD"; "GI"; "GENERAL"; "INFECTIONS"; "INJURIES"; "MUSCULOSKELETAL"; "NERVOUS"; "RENAL"; "REPRODUCTIVE SYSTEM"; "SKIN"; "SURGICAL AND MEDICAL"; "METABOLISM"; "IMMUNE".>>

#### Add following footn d of last page:

due to reconciliation discrepancies, safety database reported AE term "Endometriosis" as a SAE, - For patient # while in clinical database this AE was not recorded as an SAE.

<sup>-</sup> Arm: 1: Arm 1; 2: Arm 2; 3: Not Randomized. Relationship to study drug: NS=Not suspected, S=Suspected.

<sup>-</sup> Action taken: A0=No action taken, A1=Study drug dosage adjusted/temp. inter., A2=Study drug perm. discont. due to this AE, A3=Concomitant medication taken, A4=Non-drug therapy given, A5=Hospitalization /Prolonged hospitalization. Day is relative to the first day of treatment (day 1). \* Event occurred during the follow-up, i.e. more than 30 days after last study treatment exposure date. ^ Event occurred between patient's informed consent date and the day before first dose of study medication. @ For patient # death occurred during consent date and the day before first dose of study medication. @ For patient # AE "PHLEGMON FOOT - BIG TOE RIGHT" is reported as PT "Cellulitis" in Survival FU. For patient # the AE listing while it is reported as PT "Osteoarthritis" in the SAE listing. PT for the same AE has been wrongly decoded and reconciliation was not requiring a perfect match of the PT.

### Listing 16.2.7-2.2 Adverse events leading to study drug discontinuation – Full Analysis Set

<<Pre>rogramming note: Same shell as serious adverse events listing (listing 16.2.7-2.1) but subset on AEs marked as leading to
study drug discontinuation.>>

- Arm: 1: Arm 1; 2: Arm 2; 3: Not Randomized. Relationship to study drug: NS=Not suspected, S=Suspected
- Action taken: A0=No action taken, A1=Study drug dosage adjusted/temporarily interrupted, A2=Study drug permanently discontinued due to this AE, A3=Concomitant medication taken, A4=Non-drug therapy given, A5=Hospitalization/Prolonged hospitalization. Day is relative to the first day of treatment (day 1).
- \* event occurred during the follow-up, i.e. more than 30 days after last study treatment exposure date.
- ^ Event occurred between patient's informed consent date and the day before first dose of study medication.
- Patient # reported as disc. Ind/Cons phase due to AE "Blast Crisis"- G2, should have been reported as disc. Ind/Cons phase due to Disease Progression, progression to Blast Crisis, as per Prot.

<<Pre>rogramming note: Abbreviated system organ class to be used for the listings i.e. removing the term disorder and
conditions:

"NEOPLASMS"; "RESPIRATORY"; "BLOOD"; "GI"; "GENERAL"; "INFECTIONS"; "INJURIES"; "MUSCULOSKELETAL"; "NERVOUS"; "RENAL"; "REPRODUCTIVE SYSTEM"; "SKIN"; "SURGICAL AND MEDICAL"; "METABOLISM"; "IMMUNE".>>

#### Add following footnote at the end of last page:

- For patient # due to reconciliation discrepancies, safety database reported AE term "Endometriosis" as a SAE, while in clinical database this AE was not recorded as an SAE.

### Listing 16.2.7-2.3 Adverse events of interest – Full Analysis Set

<<Pre>rogramming note: Same shell as serious adverse events listing (listing 16.2.7-2.1) but subset on AEs marked as Adverse
Events of Interest.>>

- Arm: 1: Arm 1; 2: Arm 2; 3: Not Randomized.
- Relationship to study drug: NS=Not suspected, S=Suspected.
- Action taken: A0=No action taken, A1=Study drug dosage adjusted/temporarily interrupted, A2=Study drug permanently discontinued due to this AE, A3=Concomitant medication taken, A4=Non-drug therapy given, A5=Hospitalization/Prolonged hospitalization.
- Day is relative to the first day of treatment (day 1)
- \* Event occurred during the follow-up, i.e. more than 30 days after last study treatment exposure date.
- ^ Event occurred between patient's informed consent date and the day before first dose of study medication.

<<Pre>rogramming note: Abbreviated system organ class to be used for the listings i.e. removing the term disorder and
conditions:

"NEOPLASMS"; "RESPIRATORY"; "BLOOD"; "GI"; "GENERAL"; "INFECTIONS"; "INJURIES"; "MUSCULOSKELETAL"; "NERVOUS"; "RENAL"; "REPRODUCTIVE SYSTEM"; "SKIN"; "SURGICAL AND MEDICAL"; "METABOLISM"; "IMMUNE".>>

## Listing 16.2.7-3.1 CV risk factors, Nilotinib exposure, glucose and total cholesterol rates for patients with cardiac and vascular adverse events of interest, Full Analysis Set

| Phase | Adverse Event Verbatim/<br>Abbreviated System organ class/<br>Preferred term | Start date/<br>End date<br>of AE (dur.) | Grade/<br>Relation/<br>Action taken | Fasting glucose (unit) / Time between assessment and AE start date* | |
|---|---|---|---|---|---|
| CV risk fact<br>Values at ba | c, Center: xxx, Patient: xxx, Arm: or at baseline: Very high/High/Moseline (units): fasting glucose: ministration: First Date: DDMMMY) | oderate/Low<br>XX (xx), total | cholesterol: > | | |
| IND/CONS | Verbatim/ Ab SOCxxxxxx/<br>PTxxxxxxxxxxx | DDMMYYYY/<br>DDMMYYYY (XX) | G1/NS/A0 | xx | xx |
| TFR | Verbatim/Ab SOCxxxxxx / PTxxxxxxxxxxxx | DDMMYYYY/<br>DDMMYYYY (XX) | G2/S/A2 | xx | xx |
| RE-TRT | Verbatim/Ab SOCxxxxxx / PTxxxxxxxxxxxx | DDMMYYYY/<br>DDMMYYYY (XX) | G2/S/A2 | xx | xx |

<sup>-</sup> Arm: 1: Arm 1; 2: Arm 2; 3: Not Randomized.

<<Pre><<Pre>rogramming note: Selected AE with Abbreviated system organ class equal to 'Cardiac disorders' or 'Vascular disorders' and
CVEs not empty. Relative line of treatment and laboratory assessments should be flag with RECIN [derived.a\_ aev].
Adverse Event Verbatim/...: AEVNAM1AX/ ABBR SOC/ PT TXTX [derived.a\_ aev]

Start date of AE/ day: AEVSTT1D/ AEDAY\_1N [derived.a\_ aev]

End date of AE/ day: AEVEND1D/ AEEND 1N [derived.a aev]

AE dur: AEDUR 1N [derived.a aev]

Grade/...: AEVGRD2C/ AEVSMR2C/ ACNTAKC [derived.a aev]

Fasting glucose (unit) / Time between assessment and AE start date

Total cholesterol (unit) / Time between assessment and AE start date >>

<sup>-</sup> Phase: IND/CONS = induction/consolidation phase, TFR=treatment free remission phase and RE-TRT=re-treatment phase.

<sup>-</sup> Relationship to study drug: NS=Not suspected, S=Suspected

<sup>-</sup> Action taken: A0=No action taken, A1=Study drug dosage adjusted/temporarily interrupted, A2=Study drug permanently discontinued due to this AE, A3=Concomitant medication taken, A4=Non-drug therapy given, A5=Hospitalization/Prolonged hospitalization.

<sup>-</sup> Day is relative to the first day of treatment (day 1).

<sup>\*</sup> The last available assessment before or at date of start of the event is considered.

Novartis Confidential Page 441 RAP Module 7.1 Confidential Protocol No CAMN107AIC0

### Listing 16.2.7-3.2 Cardiac and vascular adverse events of interest, Full Analysis Set

| Phase | Adverse<br>Event<br>Abbrevia<br>ted<br>System<br>organ<br>class | Adverse<br>Event<br>Verbatim | Adverse<br>Event<br>Preferred<br>term | CVEs | Start date<br>of AE (day) | End date of AE<br>(day) | AE<br>Dur. | Grade/<br>Relation/<br>Action taken |
|---|---|---|---|---|---|---|---|---|
| Age: xxx, | Sex: xxx, F | Race: xxx | t: xxx, Arm: xx pate: DDMMMYYYY, | Last Date: DDMMMYYYY | | | | |
| IND/CONS | Ab<br>SOCxxxxx<br>x | Verbatim | PTxxxxxxxxxx | IHD/PAOD/ICE/Others | DDMMMYYYY (XX) | DDMMMYYYY (XX) | XX | G1/NS/A0 |
| | Ab<br>SOCxxxxx<br>x | Verbatim | PTxxxxxxxxxx | IHD/PAOD/ICE/Others | DDMMMYYYY (XX) | DDMMMYYYY (XX) | XX | G2/S/A2 |

<sup>-</sup> Arm: 1: Arm 1; 2: Arm 2; 3: Not Randomized.

<<Pre>rogramming note: Selected AE with Abbreviated system organ class equal to 'Cardiac disorders' or 'Vascular disorders' and
CVEs not empty

Total study period.

Treatment Administration: First Date: datepart(STTEXP10), Last Date: datepart(ENDEXP10) [derived.a dar]

Adverse Event Abbreviated System organ class: ABBR SOC [derived.a aev]

Adverse Event Verbatim: AEVNAM1AX [derived.a\_ aev]
Adverse Event Preferred term: PT TXTX [derived.a\_ aev]

CVEs: AEVSG1/ AEVSG2/ AEVSG3/AEVSG4

<sup>-</sup> Phase: IND/CONS = induction/consolidation phase, TFR=treatment free remission phase and RE-TRT=re-treatment phase.

<sup>-</sup> IHD: Ischemic heart disease, PAOD: Peripheral arterial occlusive disease, ICE: Ischemic cerebrovascular events

<sup>-</sup> Relationship to study drug: NS=Not suspected, S=Suspected

<sup>-</sup> Action taken: A0=No action taken, A1=Study drug dosage adjusted/temporarily interrupted, A2=Study drug permanently discontinued due to this AE, A3=Concomitant medication taken, A4=Non-drug therapy given, A5=Hospitalization/Prolonged hospitalization

<sup>-</sup> Day is relative to the first day of treatment (day 1).

Novartis Confidential Page 442 RAP Module 7.1 Confidential Protocol No CAMN107AIC0

Start date of AE/ day: AEVSTT1D/ AEDAY\_1N [derived.a\_ aev]
End date of AE/ day: AEVEND1D/ AEEND\_1N [derived.a\_ aev]
AE dur: AEDUR\_1N [derived.a\_ aev], Grade/...: AEVGRD2C/ AEVSMR2C/ ACNTAKC [derived.a\_ aev]>>

# Listing 16.2.7-3.3 Outcomes and subsequent concomitant medications for patients with cardiac adverse events of interest, Full Analysis Set

Concomitant medications\*

Phase Date of first First cardiac event Number of Date of study Reason for Preferred Start date (day) (cardiac event/ Verbatim/ Abbreviated discontinuatio study cardiac term/ System organ class/ events n/ day discontinuat Verbatim / on Preferred term ion

Country: xxx, Center: xxx, Patient: xxx, Arm:xx Age: xxx, Sex: xxx, Race: xxx

Treatment Administration: First Date: DDMMMYYYY, Last Date: DDMMMYYYY

Date of last contact (day): DDMMMYYYY (XX)

IND/CONS DDMMMYYYY/ XX SOCxxxxxx/ Verbatim/ XX DDMMMYYYY/ XX xxxxxx PTXXXXX/ XXXX DDMMMYYYY (XX)
PTxxxxxxxx

<sup>-</sup> Arm: 1: Arm 1; 2: Arm 2; 3: Not Randomized.

<sup>-</sup> Phase: IND/CONS = induction/consolidation phase, TFR=treatment free remission phase and RE-TRT=re-treatment phase.

<sup>-</sup> Day is relative to the first day of treatment (day 1).

<sup>- \*</sup> Concomitant medications after the date of start of the first event where the indication is related to cardiovascular diseases. If the date of start of the first event is missing or incomplete then all concomitant medications after day 1 are displayed.

## Listing 16.2.7-3.4 Outcomes and subsequent concomitant medications for patients with vascular adverse events of interest, Full Analysis Set

Concomitant medications\* Indication Phase Date of First vascular event Number of Date of study Reason for Preferred Start. first Abbreviated System organ vascular discontinuatio study term/ date (day) vascular class/ Verbatim/ events n/ dav discontinuat Verbatim / event / day Preferred term ion Country: xxx, Center: xxx, Patient: xxx, Arm: xx Age: xxx, Sex: xxx, Race: xxx Treatment Administration: First Date: DDMMMYYYY, Last Date: DDMMMYYYY Date of last contact (day): DDMMMYYYY (XX) Phase DDMMMYYYY DDMMMYYYY/ XX SOCxxxxxx/ Verbatim/ XX XXXXXX PTXXXXX/ XXXX DDMMMYYYY / XX PTxxxxxxx XXXXX (XX)

<sup>-</sup> Arm: 1: Arm 1; 2: Arm 2; 3: Not Randomized.

<sup>-</sup> Phase of the event: IND/CONS = induction/consolidation phase, TFR=Treatment free remission phase and RE-TRT=Re-treatment phase.

<sup>-</sup> Day is relative to the first day of each phase (day 1)

<sup>- \*</sup> Concomitant medications after the date of start of the first event where the indication is related to cardiovascular diseases. If the date of start of the first event is missing or incomplete then all concomitant medications after day 1 are displayed.

### **Section 16.2.8 – Laboratory measurements**

### Listing 16.2.8-1.1 Hematology laboratory values and normal ranges – Full Analysis Set

| Country/ Center/<br>Patient/ Arm | Age/<br>Sex/<br>Race | Phase/ Sample<br>date/ Day | Test | Value<br>(SI Unit) | Normal<br>Range | Grade |
|---|---|---|---|---|---|---|
| XXX/0XXX/0XXXX/X | XX/X/XX | IND/CONS1/CONS2/<br>TFR/RE-TRT<br>DDMMMYYYY/XX | Hemoglobin | XX (LB/%) | L/N/H | Gx |
| | | | Platelets | XX (LB/%) | L/N/H | Gx |
| | | | WBC | XX (LB/%) | L/N/H | Gx |
| | | | Absolute Neutrophils/ Neutrophils | XX (LB/%) | L/N/H | Gx |
| | | | Absolute Lymphocytes/ Lymphocytes | XX (LB/%) | L/N/H | Gx |
| | | | Absolute Eosinophils/ Eosinophils | XX (LB/%) | L/N/H | |
| | | | Absolute Basophils/ Basophils | XX (LB/%) | L/N/H | |
| | | | Absolute Monocytes/ Monocytes | XX (LB/%) | L/N/H | |
| | | | Absolute Promyelocytes/ Promyelocytes | XX (LB/%) | L/N/H | |
| | | | Absolute Myelocytes/ Myelocytes | XX (LB/%) | L/N/H | |
| | | | Absolute Metamyelocytes/ Metamyelocytes | XX (LB/%) | L/N/H | |
| | | | Absolute Blasts/ Blasts | XX (LB/%) | L/N/H | |
| | | | Absolute Other/ Other | | | |
| | | | XXX | XX (LB/%) | L/N/H | Gx |

<sup>-</sup> Arm: 1: Arm 1; 2: Arm 2; 3: Not Randomized.

"Note for programming: When absolute and percentage value are provided, given both Grade are to display only for laboratory tests where CTCAE grades are defined"

<sup>-</sup> M: Male; F: Female; W: White; B: Black or African American; A: Asian; AI: American Indian or Alaska Native; N: Native Hawaiian or other Pacific Islander; UK: Unknown; O: Other.

<sup>-</sup> Phase: IND=ind. phase (0-12 months), CONS1 = pre-rand. cons. phase (12-24 months), CONS2 = post-rand. cons. phase (ARM 2) (24-36 months), TFR=treatment free remission phase and RE-TRT=re-treatment phase.

<sup>-</sup> L/H denotes a value below/above normal range, N denotes normal.

<sup>-</sup> Gx denotes an abnormal high value meeting toxicity CTCAE grading criteria and G-x an abnormal low value according to toxicity CTCAE grading. Day is relative to the first day of treatment (day 1).

## Listing 16.2.8-2.1 Biochemistry laboratory values and normal ranges – Full Analysis Set

| | | ioti y laborator y | valace and normal ranges | i an maryolo cot | | |
|---|---|---|---|---|---|---|
| Country/<br>Center/<br>Patient/ Arm | Age/<br>Sex/<br>Race | Phase/ Sample<br>date/ Day | Test | Value<br>(SI Unit) | Normal<br>Range | Grade |
| XXX/0XXX/0XXXX/<br>X | XX/X/XX | IND/CONS1/<br>CONS2/TFR/RE-<br>TRT<br>DDMMMYYYY/XX | Creatine | XX (LB/%) | L/N/H | Gx |
| | | | Hypoglycemia | XX (LB/%) | L/N/H | Gx |
| | | | Hyperglycemia | XX (LB/%) | L/N/H | Gx |
| | | | Total Cholesterol | XX (LB/%) | L/N/H | Gx |
| | | | HDL | XX (LB) | L/N/H | |
| | | | LDL | XX (LB) | L/N/H | |
| | | | Triglycerides | XX (LB/%) | L/N/H | Gx |
| | | | Total bilirubin | XX (LB/%) | L/N/H | Gx |
| | | | Direct bilirubin | XX (LB/%) | L/N/H | Gx |
| | | | Indirect bilirubin | XX (LB/%) | L/N/H | Gx |
| | | | AST/SGOT | XX (LB/%) | L/N/H | Gx |
| | | | ALT/SGPT | XX (LB/%) | L/N/H | Gx |
| | | | LDH | XX (LB) | L/N/H | |
| | | | Hyponatremia | XX (LB/%) | L/N/H | Gx |
| | | | Hypernatremia | XX (LB/%) | L/N/H | Gx |
| | | | Hypocalcemia | XX (LB/%) | L/N/H | Gx |
| | | | Hypercalcemia | XX (LB/%) | L/N/H | Gx |
| | | | Hypokalemia | XX (LB/%) | L/N/H | Gx |
| | | | Hyperkalemia | XX (LB/%) | L/N/H | Gx |
| | | | Hypomagnesemia | XX (LB/%) | L/N/H | Gx |
| | | | Hypermagnesemia | XX (LB/%) | L/N/H | Gx |
| | | | Phosphorus | XX (LB/%) | L/N/H | Gx |
| | | | Lipase | XX (LB/%) | L/N/H | Gx |

| Novartis<br>RAP Module 7.1 | Confidential<br>6-May-2021 (14:35) | | Page 447<br>Protocol No CAMN107AIC0 | |
|---|---|---|---|---|
| | Amylase | XX (LB/%) | L/N/H | Gx |
| | HbA1C | XX (LB) | L/N/H | |
| | Alkaline Phosphatase Increase | XX (LB/%) | L/N/H | Gx |
| | Hypoalbuminemia | XX (LB/%) | L/N/H | Gx |

<sup>-</sup> Arm: 1: Arm 1; 2: Arm 2; 3: Not Randomized.

 $\verb§`Note for programming: Grade will be display only for laboratory tests where CTCAE grades are defined"$ 

<sup>-</sup> M: Male; F: Female; W: White; B: Black or African American; A: Asian; AI: American Indian or Alaska Native; N: Native Hawaiian or other Pacific Islander; UK: Unknown; O: Other.

<sup>-</sup> Phase: IND = ind. phase (0-12 months), CONS1 = pre-rand. cons., CONS2 = post-rand.n cons. phase (ARM 2) (24-36 months), TFR=treatment free remission phase, RE-TRT=re-treatment phase.

<sup>-</sup> L/H denotes a value below/above normal range, N denotes normal range.

<sup>-</sup> Gx denotes an abnormal high value meeting toxicity CTCAE grading criteria and G-x an abnormal low value according to toxicity CTCAE grading. Day is relative to the first day of treatment (day 1).

## Listing 16.2.8-3.1 Hematological data and molecular response in patients with absolute blasts higher than normal ranges, Full Analysis Set

| | Phase/<br>Time-Windows/<br>Visit/<br>Date of visit | %<br>Blasts<br>(range) | | % Promye locytes (range) | %<br>Basophils<br>(range) | %<br>Myelocytes<br>(range) | % Meta- myelocytes (range) | Platelets<br>10E9/L | WBC<br>10E9/L | %<br>BCR-ABL<br>/ABL<br>(IS) | Derived<br>MR | Derived<br>loss of<br>MMR or<br>MR 4.0 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| , | ARM: x, Countr | - | • | | | • | ace: xxx | | | | | _ |
| | Treatment Admi | .nistration: | First Date: | : DDMMMYYY | Y, Last Date | e: DDMMMYYYY | | | | | | |
| | IND /M3/V1-M3<br>/DDMMMYYYY | XX<br>(L/N/H) | XX | XX<br>(L/N/H) | XX<br>(L/N/H) | XX<br>(L/N/H) | XX<br>(L/N/H) | XX | XX | XX | <3 | |
| | IND/M6/UNSCH<br>/DDMMMYYYY | XX<br>(L/N/H) | XX | XX<br>(L/N/H) | XX<br>(L/N/H) | XX<br>(L/N/H) | XX<br>(L/N/H) | XX | XX | XX | 4.5 | |
| | TFR/M6/UNSCH<br>/DDMMMYYYY | XX<br>(L/N/H) | XX | XX<br>(L/N/H) | XX<br>(L/N/H) | XX<br>(L/N/H) | XX<br>(L/N/H) | XX | XX | XX | <3 | Loss of<br>MMR |

<sup>-</sup> Arm: 1: Arm 1; 2: Arm 2; 3: Not Randomized.

<< Programming note: For each patient merge PCR data with haematological data by time-point and visit. If there are several unscheduled visits in a same time-window then merge them by incremental order defined by chronology >>

<sup>-</sup> L/N/H denotes categories defined by normal ranges.

<sup>-</sup> BASE=Baseline; SCR=Screening; RANDO = Randomization; EOP = End Of Phase; UNSCH = Unscheduled visit; IND = induction phase (0-12 months), CONS1 = pre-randomization consolidation phase, CONS2 = post-randomization consolidation phase (ARM 2)(24-36 months), TFR=Treatment free remission phase and RE-TRT=Re-treatment phase. - PCR assessments, laboratory assessments and bone marrow assessments are merged together by visit number, visit date and visit name.

<sup>-</sup> When patients are in molecular response 4.5 then Molecular Response (MR) is equal to 4.5, if patients are in molecular response 4.0 then MR is equal to 4, if patients are in major molecular response then MR is equal to 3, if none of those responses are defined but BCR-ABL (IS) ratio > 0.1 then MR is equal to <3.

## Listing 16.2.8-3.2 Hematological data and molecular response in patients with absolute metamyelocytes higher than normal ranges, Full Analysis Set

| Phase<br>Time<br>Winde<br>/<br>Visi | - (range)<br>ows | %<br>Blasts<br>in bone<br>marrow | <pre>% Promye Locytes (range)</pre> | %<br>Basophils<br>(range) | %<br>Myelocytes<br>(range) | %<br>Metamyelocytes<br>(range) | Platelets<br>10E9/L | WBC<br>10E9/L | % BCR-<br>ABL/ABL<br>(IS) | Molecular<br>Response<br>Derived |
|---|---|---|---|---|---|---|---|---|---|---|
| ARM:<br>xxx<br>Trea | - | · | | · | Age: xxx, Sex Last Date: DI | x: xxx, Race: | | | | |
| M3/<br>V1-N | XX<br>I3 (L/N/H) | XX | XX<br>(L/N/H) | XX<br>(L/N/H) | XX (L/N/H) | XX (L/N/H) | XX | XX | XX | <3 |
| M6/<br>UNSO | XX<br>H (L/N/H) | XX | XX<br>(L/N/H) | XX<br>(L/N/H) | XX (L/N/H) | XX (L/N/H) | XX | XX | XX | 4.5 |

<sup>-</sup> Arm: 1: Arm 1; 2: Arm 2; 3: Not Randomized.

<<Pre>rogramming note: For each patient merge PCR data with haematological data by time-point and visit. If there are several
unscheduled visit in a time-window then merge them by incremental order defined by chronology >>

<sup>-</sup> L/N/H denotes categories defined by normal ranges

<sup>-</sup> BASE=Baseline; SCR=Screening; RANDO = Randomization; EOP = End Of Phase; UNSCH = Unscheduled visit; IND = induction phase (0-12 months), CONS1 = pre-randomization consolidation phase (0-24 months), CONS2 = post-randomization consolidation phase (ARM 2) (24-36 months), TFR=Treatment free remission phase and RE-TRT=Re-treatment phase.

<sup>-</sup> PCR assessments, laboratory assessments and bone marrow assessments are merged together by visit number, visit date and visit name

<sup>-</sup> When patients are in molecular response 4.5 then Molecular Response is equal to 4.5, if patients are in molecular response 4.0 then Molecular Response is equal to 4, if patients are in major molecular response then Molecular Response is equal to 3, if none of those responses are defined but BCR-ABL (IS) ratio > 0.1 then Molecular Response is equal to <3.

### Section 16.2.9 – Vital signs, physical findings and other observations related to safety listings

### Listing 16.2.9-1.1 Vital signs – Full Analysis Set

| Country/ Center/<br>Patient/ Arm | Age/Sex/Race | Cardiovascular<br>Event (type) | Visit | Weight<br>(kg) | Body<br>temperature<br>(C) | Sitting<br>Pulse<br>(bpm) | Sitting Blood pressure Systolic/Diastolic (mmHg) |
|---|---|---|---|---|---|---|---|
| XXX/0XXX/0XXXX/1 | XX/X/XX | Yes (IHD, ICE) | Screening | XX.X | XX.X | XX | XX.X / XX.X |
| | | | Month 3 | XX.X | XX.X | XX | XX.X / XX.X |
| | | | Month 6 | XX.X | XX.X | XX | XX.X / XX.X |
| | | | Month 9 | XX.X | XX.X | XX | XX.X / XX.X |
| | | | | | | | ••• |
| | | | Month 24 | XX.X | XX.X | XX | XX.X / XX.X |
| XXX/0XXX/0XXXX/2 | XX/X/XX | No | Screening | XX.X | XX.X | XX | XX.X / XX.X |
| | | | • • • | • • • | • • • | • • • | • • • |
| | | | Month 24 | XX.X | XX.X | XX | XX.X / XX.X |
| | | | • • • | | | • • • | ••• |
| | | | Month 36 | XX.X | XX.X | XX | XX.X / XX.X |

<sup>-</sup> Arm: 1: Arm 1; 2: Arm 2; 3: Not Randomized.

<sup>-</sup> M: Male; F: Female; W: White; B: Black or African American; A: Asian; AI: American Indian or Alaska Native; N: Native Hawaiian or other Pacific Islander; UK: Unknown; O: Other.

<sup>-</sup>CVE categories: IHD: Ischemic heart disease, PAOD: Peripheral arterial occlusive disease, ICE: Ischemic cerebrovascular events), Others.

### Listing 16.2.9-2.1 Electrocardiograms – Full Analysis Set

| Country/ Center/<br>Patient/ Arm | Age/Sex/Race | Phase | Date of ECG | QTcF interval (msec) | Clinically significant abnormalities present? | If clinically significant, specify |
|---|---|---|---|---|---|---|
| XXX/0XXX/0XXXX/X | XX/X/XX | IC | DDMMMYYYY | XX | Yes/No | XXXXXXXX |
| | | IC | DDMMMYYYY | XX | Yes/No | XXXXXXXX |
| Repea | nt for each asse | essment | | | | |
| XXX/0XXX/0XXXX/X | XX/X/XX | IC | DDMMMYYYY | XX | Yes/No | XXXXXXXX |
| | | IC | DDMMMYYYY | XX | Yes/No | XXXXXXXX |
| Repea | nt for each asse | essment | | | | |

<sup>-</sup> Arm: 1: Arm 1; 2: Arm 2; 3: Not Randomized.

### **Listing 16.2.9-2.2 Echocardiography – Full Analysis Set**

| Country/ Center/<br>Patient/ Arm | Age/Sex/Race | Phase | Date of<br>Echocardiography | LVEF | Interpretation | If clinically significant, specify |
|---|---|---|---|---|---|---|
| XXX/0XXX/0XXXX/X | XX/X/XX | IC | DDMMMYYYY | XX | N/CI/CS | XXXXXXXX |
| | | IC | DDMMMYYYY | XX | N/CI/CS | XXXXXXXX |
| | Repeat for each as | ssessment | | | | |
| XXX/0XXX/0XXXX/X | XX/X/XX | IC | DDMMMYYYY | XX | N/CI/CS | XXXXXXXX |
| | | IC | DDMMMYYYY | XX | N/CI/CS | XXXXXXXX |
| | Repeat for each as | ssessment | | | | |

<sup>-</sup> Arm: 1: Arm 1; 2: Arm 2; 3: Not Randomized.

<sup>-</sup> M: Male; F: Female; W: White; B: Black or African American; A: Asian; AI: American Indian or Alaska Native; N: Native Hawaiian or other Pacific Islander; UK: Unknown; O: Other.

<sup>-</sup> Phase: IND = induction phase (0-12 months), CONS1 = pre-randomization consolidation phase (0-24 months), CONS2 = post-randomization consolidation phase (ARM 2) (24-36 months), TFR=treatment free remission phase and RE-TRT=re-treatment phase.

<sup>-</sup> M: Male; F: Female; W: White; B: Black or African American; A: Asian; AI: American Indian or Alaska Native; N: Native Hawaiian or other Pacific Islander; UK: Unknown; O: Other.
ND: Not Done.

<sup>-</sup> Phase: IND = induction phase (0-12 months), CONS1 = pre-randomization consolidation phase (0-24 months), CONS2 = post-randomization consolidation phase (ARM 2) (24-36 months), TFR=treatment free remission phase and RE-TRT=re-treatment phase.

<sup>-</sup> Interpretation: N=Normal, CI=Clinically insignificant abnormality, CS=Clinically significant abnormality.

### Listing 16.2.9-3.1 Concomitant medications – Full Analysis Set

| Country/<br>Center/<br>Patient/ Arm | Age/ Sex/<br>Race | Preferred<br>term/ Verbatim | ATC<br>level 2 | Indication | Start/End<br>dates | Phase | Route of administration | Dose (units)/<br>Frequency |
|---|---|---|---|---|---|---|---|---|
| XXX/0XXX/0XXXX<br>/X | XX/X/XX | PTXXXXX/XXXXX | XXXXX | XXXXX | DDMMMYYYY<br>/<br>DDMMMYYYY | IND | XXXXX | XX (X) / XX |
| XXX/0XXX/0XXXX<br>/X | XX/X/XX | PTXXXXX/XXXXX | XXXXX | XXXXX | DDMMMYYYY<br>/<br>DDMMMYYYY | RE-TRT | XXXXX | XX (X) / XX |

<sup>-</sup> Arm: 1: Arm 1; 2: Arm 2; 3: Not Randomized.

### Listing 16.2.9- 3.2 Prohibited concomitant medications – Full Analysis Set

| Country/<br>Center/<br>Patient/ Arm | Age/ Sex/<br>Race | Preferred<br>term/ Verbatim | ATC<br>level 2 | Indication | Start/End<br>dates | Phase | Route of administration | Dose (units)/<br>Frequency |
|---|---|---|---|---|---|---|---|---|
| XXX/0XXX/0XXXX<br>/X | XX/X/XX | PTXXXXX/XXXXX | XXXXX | XXXXX | DDMMMYYYY<br>/<br>DDMMMYYYY | CONS1 | XXXXX | XX (X) / XX |
| XXX/0XXX/0XXXX<br>/X | XX/X/XX | PTXXXXX/XXXXX | XXXXX | XXXXX | DDMMMYYYY<br>/<br>DDMMMYYYY | CONS2 | XXXXX | XX (X) / XX |

<sup>-</sup> Arm: 1: Arm 1; 2: Arm 2; 3: Not Randomized.

<sup>-</sup> M: Male; F: Female; W: White; B: Black or African American; A: Asian; AI: American Indian or Alaska Native; N: Native Hawaiian or other Pacific Islander; UK: Unknown; O: Other.

<sup>-</sup> Phase: IND = induction phase, CONS1 = pre-randomization consolidation phase (0-24 months, CONS2 = post-randomization consolidation phase (ARM 2) (24-36 months), TFR=treatment free remission phase and RE-TRT=re-treatment phase.

<sup>-</sup> M: Male; F: Female; W: White; B: Black or African American; A: Asian; AI: American Indian or Alaska Native; N: Native Hawaiian or other Pacific Islander; UK: Unknown; O: Other.

<sup>-</sup> Phase: CONS1 = pre-randomization consolidation phase (0-24 months, CONS2 = post-randomization consolidation phase (ARM 2) (24-36 months).

### Listing 16.2.9-4.1 Prior Imatinib therapy— Full Analysis Set

| Country/<br>Center/<br>Patient/ Arm | Age/ Sex/<br>Race | Start/End<br>dates | Route of administration | Dose (units)/<br>Frequency | Therapy<br>type | Reason for discontinuat ion |
|---|---|---|---|---|---|---|
| XXX/0XXX/0XXXX<br>/X | XX/X/XX | DDMMMYYYY/<br>DDMMMYYYY | XXXXX | XX (X) / XX | Chemotherapy | xxxxxxxxx |
| XXX/0XXX/0XXXX<br>/X | XX/X/XX | DDMMMYYYY/<br>DDMMMYYYY | XXXXX | XX (X) / XX | Targeted<br>therapy | xxxxxxxxxx |

<sup>-</sup> Arm: 1: Arm 1; 2: Arm 2; 3: Not Randomized.

### Listing 16.2.9-4.2 Prior antineoplastic therapy, other than Imatinib – Full Analysis Set

| Country/<br>Center/<br>Patient/ Arm | Age/ Sex/<br>Race | Preferred<br>term/<br>Verbatim | ATC<br>level<br>2 | Start/End<br>dates | Route of administ ration | Dose (units)/<br>Frequency | Therapy<br>type | Reason for discontinuation |
|---|---|---|---|---|---|---|---|---|
| XXX/0XXX/0XXX<br>X/X | XX/X/XX | PTXXXXX/XXXXX | XXXXX | DDMMMYYYY/<br>DDMMMYYYY | XXXXX | XX (X) / XX | Chemotherapy | xxxxxxxxx |
| XXX/0XXX/0XXX<br>X/X | XX/X/XX | PTXXXXX/XXXXX | XXXXX | DDMMMYYYY/<br>DDMMMYYYY | XXXXX | XX (X) / XX | Targeted<br>therapy | xxxxxxxxxx |

<sup>-</sup> Arm: 1: Arm 1; 2: Arm 2; 3: Not Randomized.

<sup>-</sup> M: Male; F: Female; W: White; B: Black or African American; A: Asian; AI: American Indian or Alaska Native; N: Native Hawaiian or other Pacific Islander; UK: Unknown; O: Other.

<sup>-</sup> M: Male; F: Female; W: White; B: Black or African American; A: Asian; AI: American Indian or Alaska Native; N: Native Hawaiian or other Pacific Islander; UK: Unknown; O: Other.

| <b>Listing 16.2.9-5.1</b> | Survival follow-up- Full Analysis se | et |
|---------------------------|--------------------------------------|----|
|---------------------------|--------------------------------------|----|

| | | | | | If no | | If yes<br>or Lost<br>to<br>follow-<br>up | | | If rece<br>any<br>treat | TKI |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Country/<br>Center/<br>Patient/<br>Arm | Age/<br>Sex/<br>Race | Visit | Is the<br>Subjec<br>t<br>alive | Date<br>of<br>death | Princip<br>al<br>cause<br>of<br>Death | If<br>other<br>speci<br>fy | Last<br>date<br>of<br>contact<br>? | Did patient undergo stem-cell transplant / Is the disease progressing to AP/BP ? | Is the patient receivi ng any TKI treatme nt ? | Treatment | If<br>other<br>specify |
| XXX/0XXX/<br>0XXXX/X | XX/X/<br>XX | FU-Month | Yes | | | | | Yes/No | Yes | Nilotinib | |
| XXX/0XXX/<br>0XXXX/X | XX/X/<br>XX | FU-Month<br>6 | Yes | | | | DDMMMYY<br>YY | Yes/No | No | | |
| XXX/0XXX/<br>0XXXX/X@ | XX/X/<br>XX | FU-Month<br>36 | Yes | | | | DDMMMYY<br>YY | Yes/No | Yes | Other | xxxxxx |
| XXX/0XXX/<br>0XXXX/X | XX/X/<br>XX | FU-Month<br>3 | No | DDMMMYYYY | Study<br>indicat<br>ion<br>(CML) | | | | | | |
| <br>XXX/0XXX/<br>0XXXX/X | XX/X/<br>XX | FU-Month<br>3 | No | DDMMMYYYY | Other | XXXXX | | | | | |

<sup>-</sup> Arm: 1: Arm 1; 2: Arm 2; 3: Not Randomized.

<sup>-</sup> M: Male; F: Female; W: White; B: Black or African American; A: Asian; AI: American Indian or Alaska Native; N: Native Hawaiian or other Pacific Islander; UK: Unknown; O: Other.

<sup>@</sup> For patient # death occurred during Survival follow-up.

## Listing 16.2.9-5.2 Safety follow-up- Full Analysis set

| Country/ Center/<br>Patient/ Arm | Age/<br>Sex/<br>Race | Safety follow<br>up performed | Date of<br>clinical<br>visit/<br>telephone<br>call | In case of telephone call Medical intervention necessary? | Date of<br>Medical<br>intervention | Reason for<br>safety<br>follow up<br>Not Performed |
|---|---|---|---|---|---|---|
| XXX/0XXX/0XXXX/X | XX/X/XX | During Clinical visit | DDMMMYYYY | | | |
| XXX/0XXX/0XXXX/X@ | XX/X/XX | During Telephone call | DDMMMYYYY | Yes | DDMMMYYYY | |
| XXX/0XXX/0XXXX/X | XX/X/XX | No | | | | xxxxxxxxxx |

<sup>-</sup> Arm: 1: Arm 1; 2: Arm 2; 3: Not Randomized.

<sup>-</sup> M: Male; F: Female; W: White; B: Black or African American; A: Asian; AI: American Indian or Alaska Native; N: Native Hawaiian or other Pacific Islander; UK: Unknown; O: Other.

<sup>@</sup> For patient # death occurred during Survival follow-up.

### Listing 16.2.9-6 Prior imatinib exposure – LSC sub-study Full Analysis Set

| Country/<br>Center/<br>Patient/<br>Arm | Age/<br>Sex/<br>Race | Prior<br>Imatinib<br>intake | Duration<br>of prior<br>exposure<br>(months) | Duration of prior exposure category (years) | Sokal<br>Score<br>at<br>diagnosis | Sokal<br>Score category<br>at<br>diagnosis |
|---|---|---|---|---|---|---|
| XXX/0XXX/0XXXX/X | XX/X/XX | YES | xx.x | <2 | xx.x | Low risk |
| XXX/0XXX/0XXXX/X | XX/X/XX | NO | XX.X | | XX.X | Low risk |
| XXX/0XXX/0XXXX/X | XX/X/XX | YES | xx.x | >=2 - <5 | xx.x | High risk |
| XXX/0XXX/0XXXX/X | XX/X/XX | YES | XX.X | >=5 | xx.x | Intermediate risk |

<sup>1:</sup> ARM 1; 2: ARM 2; 3: Not Randomized. M: Male; F: Female;

W: White; B: Black or African American; A: Asian; AI: American Indian or Alaska Native; N: Native Hawaiian or other Pacific Islander; UK: Unknown; O: Other.

Sokal score category: low risk (<0.8), intermediate risk (>=0.8-<=1.2) and high risk (>1.2).